

# Clinical Study Protocol 747-209 OBETICHOLIC ACID

A Phase 2, Randomized, Double-Blind, Placebo-Controlled Clinical Study Investigating the Effects of Obeticholic Acid and Atorvastatin Treatment on Lipoprotein Metabolism in Subjects with Nonalcoholic Steatohepatitis

# The CONTROL Study <u>Combination OCA aNd STatins for MonitoRing Of Lipids</u>

Version 4: 19 December 2016

# **Sponsor**

Intercept Pharmaceuticals, Inc. 4760 Eastgate Mall San Diego, CA 92121

USA

TEL: +1 858 652 6800

FAX: +1 858 558 5961

#### **CONFIDENTIAL**

The information contained herein is the property of Intercept Pharmaceuticals, Inc. and may not be reproduced, published, or disclosed to others without written authorization of Intercept Pharmaceuticals, Inc.

# SPONSOR'S APPROVAL OF THE PROTOCOL

Reviewed and Approved by:

Leigh MacConell, PhD

Vice President, Clinical Development Intercept Pharmaceuticals, Inc.

----

Date

## **INVESTIGATOR'S AGREEMENT**

I have received and read the current version of the Investigator's Brochure (IB) for obeticholic acid (OCA) and this Protocol 747-209. Having fully considered all the information available, I agree that it is ethically justifiable to give OCA to selected subjects according to this protocol.

I understand that all information concerning OCA supplied to me by the Sponsor, Intercept Pharmaceuticals, Inc., and/or its agents in connection with this study and not previously published is confidential information. This includes the IB, clinical study protocol, electronic case report forms (eCRFs), and any other preclinical and clinical data provided by the Sponsor.

I understand that no data are to be made public or published without prior knowledge and written approval by the Sponsor.

By my signature below, I hereby attest that I have read, understood and agreed to abide by all the conditions, instructions and restrictions contained in Protocol 747-209 and in accordance with Good Clinical Practice (CPMP/ICH/135/95), the Declaration of Helsinki and all regulatory requirements for protection of human subjects in clinical studies and privacy requirements for the protection of individual and company data.

I acknowledge that the Sponsor of the study has the right to discontinue the study at any time.

| Investigator's Name (Printed) | |
|-------------------------------|------|
| Investigator's Signature | Date |

#### STUDY PERSONNEL CONTACT INFORMATION

#### **Medical Monitor**

Investigators are encouraged to call the PRA Medical Support Center phone number for the United States and Canada at +1 866 326 5053 or send an email to the NASH medical monitor at CONTROL@prahs.com with safety questions as these lines of contact are monitored 24 hours a day.

Primary Medical Monitor Emad Basta, MD

Contact: (Lead) Medical Monitor/Medical Expert

PRA Health Sciences

Phone: +1 866 326 5053

Email CONTROL@prahs.com

Secondary Contact: Tolga Baykal, MD, PhD

Medical Director, Clinical Development Intercept Pharmaceuticals, Inc. (Intercept)

Mobile Phone: +1 619 643 8886 (Pacific time zone)
Email tolga.baykal@interceptpharma.com

Secondary Contact: Barbara Scholz, MD,

Medical Director, Drug Safety

Intercept

Mobile Phone: +1 858 353 1350 (Pacific time zone)
Email: barbara.scholz@interceptpharma.com

# **Clinical Operations and Project Management**

Contact: Shawn Sheeron

**Executive Director, Clinical Operations** 

Intercept

Telephone: + 1 858 964 1572 (Pacific time zone)

Mobile: + 1 215 796 3286 Fax: + 1 858 558 5961

Email: ssheeron@interceptpharma.com

#### 2. SYNOPSIS

#### Name of Sponsor/Company:

Intercept Pharmaceuticals, Inc.

#### Name of Investigational Product:

Obeticholic Acid

#### Name of Active Ingredient:

Obeticholic Acid (OCA); 6α-ethyl-chenodeoxycholic acid (6-ECDCA); INT-747; DSP-1747

#### Title of Study:

A Phase 2, Randomized, Double-Blind, Placebo-Controlled Clinical Study Investigating the Effects of Obeticholic Acid and Atorvastatin Treatment on Lipoprotein Metabolism in Subjects with Nonalcoholic Steatohepatitis

#### **Study Center(s):**

Approximately 30 investigational sites in the United States

| Study Period: | Phase of Development: |
|---|---|
| Duration of individual subject participation: up to 5 weeks in Screening (depend | ing Phase 2 |
| on current statin use) and 16 weeks during the double-blind treatment phase, | |
| followed by an optional open-label long-term safety extension (LTSE) expected | to |
| last approximately 2 years. | |

#### **Objectives:**

#### Primary Objective

• To evaluate the effect of OCA on low-density lipoprotein (LDL) metabolism in subjects with biopsy-confirmed nonalcoholic steatohepatitis (NASH) and to assess the ability of atorvastatin to modulate this effect

#### Secondary Objectives

- To evaluate the safety and tolerability of OCA alone and in combination with atorvastatin therapy in subjects with biopsy-confirmed NASH
- To evaluate the effect of OCA, with and without atorvastatin therapy, on
  - High-density lipoprotein (HDL), very low-density lipoprotein (VLDL), triglycerides (TGs), total cholesterol, and apolipoprotein concentrations
  - Components of the reverse cholesterol transport pathway

#### **Exploratory Objectives**

- To evaluate the effect of OCA on
  - Liver biochemistry, inflammation, and apoptosis
  - Markers of glucose metabolism including C-peptide, insulin, fasting plasma glucose, hemoglobin-specific A1c fraction (HbA1c), homeostatic model assessment—beta-cell function (HOMA-β) and homeostatic model assessment insulin resistance (HOMA-IR)
  - Anthropometric measures including height (measured at Screening Visit 1 only), weight, and waist and hip circumference measurements; and body mass index (BMI), and waist-to-hip ratio calculations
  - Cardiovascular risk scores (eg., Framingham Risk Score [FRS] and Reynolds score)
- To evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of OCA and its conjugates
- To evaluate the bioanalytical concentrations of atorvastatin and its metabolites
- To evaluate improvement in noninvasive-radiological assessment of fibrosis via transient elastography (TE; at sites where available)

#### Methodology:

This Phase 2, double-blind, randomized, placebo-controlled, multicenter study, with an open-label LTSE, will evaluate the effect of OCA, and the subsequent addition of statin therapy, on lipoprotein metabolism in subjects with NASH with fibrosis stage 1 to 4, but no evidence of hepatic decompensation. Approximately 80 subjects with histological evidence of definite or probable NASH, who meet all inclusion and none of the exclusion criteria will be enrolled. The histological evidence of definite or probable NASH will be based on the central reading of a liver biopsy obtained no more than 1 year prior to randomization and a nonalcoholic fatty liver disease activity score (NAS) of 4 or greater. Subjects not using statin therapy (ie, statin-free) and statin-treated subjects may be enrolled in the study. Statin-treated subjects will be required to stop statin treatment (after signing informed consent) for up to 5 weeks, including a 4-week washout period, prior to Randomization/Day 1.

#### Screening Period:

Subjects will have a screening period of up to 5 weeks prior to Randomization/Day 1.

Subjects using statins within 30 days of the initial Screening visit (Screening Visit 1) are required to stop statin therapy immediately following this initial visit and must undergo a 4-week statin washout period prior to Screening Visit 2. At Screening Visit 2, these subjects will have a pre-randomization visit for assessment of their fasting LDL cholesterol levels. Subjects with fasting LDL cholesterol values >200 mg/dL at Screening Visit 2 will be excluded from the study and their dyslipidemia should be managed according to standard of care.

Subjects who are not using statin therapy at Screening Visit 1 are required to provide a fasting blood sample at Screening Visit 2, which can occur at any time prior to randomization but after signing of the ICF. Statin-free subjects with fasting LDL cholesterol values >200 mg/dL at either Screening Visit will be excluded from the study and should be managed according to standard of care.

#### Double-Blind Phase:

At the Randomization (Day 1) Visit, subjects will be randomized in a 1:1:1:1 ratio to receive OCA 5 mg, OCA 10 mg, OCA 25 mg or placebo, orally once daily, for 16 weeks. Randomization will be stratified by LDL concentration (fasting serum LDL cholesterol at Screening Visit 2; ≤125 mg/dL or >125 mg/dL) and baseline fibrosis stage (stage 1, 2 or stage 3, 4).

At the Week 4 Visit, all subjects will initiate treatment with atorvastatin at a dose of 10 mg once daily. At the Week 8 Visit, atorvastatin will be increased to 20 mg once daily (if 10 mg daily is tolerated), and continued for an additional 4 weeks. After 4 weeks of treatment at 20 mg, the atorvastatin dose may be titrated (up or down) as clinically indicated. The final visit during the double-blind phase will occur at Week 16, after which subjects may continue into the open-label LTSE phase.

Subjects who discontinue investigational product or atorvastatin during the double-blind phase are still expected to attend scheduled study visits and are to be followed through the Week 16 Visit.

Subjects who discontinue atorvastatin during the double-blind phase are eligible to continue OCA during the double-blind phase and enroll into the LTSE at the discretion of the Investigator, provided they continue to meet the LDLc cutoff of exclusion criteria #4 (ie, LDLc <200 mg/dL).

#### LTSE Phase:

During the LTSE phase, all subjects will be treated with open-label OCA 10 mg or OCA 25 mg. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will be randomized in a 1:1 ratio to receive OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg or OCA 25 mg during the double-blind phase will continue on the same dose throughout the LTSE. During the LTSE, subjects may continue with atorvastatin therapy as clinically indicated.



LTSE = long-term safety extension; Wk = week

Note: Statin therapy refers to atorvastatin.

 $\Delta$  = Telephone safety contact at Week 6, Week 10, and Week 14

#### **Number of Subjects (Planned):**

Approximately 80 subjects with biopsy-confirmed NASH and evidence of liver fibrosis, but no hepatic decompensation, who meet eligibility criteria, will be randomized in a 1:1:1:1 ratio to 1 of 4 treatment groups. A maximum of 30% of subjects will have stage 4 fibrosis.

#### Diagnosis and Main Criteria for Inclusion:

#### **Inclusion Criteria**

Subjects must satisfy all of the following criteria to be eligible for enrollment:

- 1. Age  $\geq$ 18 years of age
- 2. Histologic evidence of NASH as assessed by central reading of a liver biopsy obtained no more than 1 year prior to randomization defined by the presence of all 3 key histological features of NASH with a score of at least 1 for each and a combined score of 4 or greater out of a possible 8 points according to NASH Clinical Research Network (CRN) criteria.
- 3. Histologic evidence of fibrosis stage 1 to stage 4 (as defined by the NASH CRN scoring of fibrosis) without any evidence of hepatic decompensation.
- 4. If subject has type 2 diabetes, is on stable dose of anti-diabetic medication (except thiazolidinediones [TZDs]) for ≥3 months prior to Day 1.
- 5. Is either not taking or is on stable doses of TZDs and/or Vitamin E for ≥6 months prior to Day 1
- 6. Contraception: Female subjects of childbearing potential must use ≥1 effective method of contraception during the study and until 30 days following the last dose of investigational product. Effective methods of contraception are considered to be those listed below.

- Barrier method, ie, condom (male or female) with spermicide or diaphragm with spermicide
- Intrauterine device
- Vasectomy (partner)
- Hormonal (eg, contraceptive pill, patch, intramuscular implant or injection)
- Abstinence (defined as refraining from heterosexual intercourse)
- 7. Must provide written informed consent and agree to comply with the study protocol including adherence to protocol-described statin withdrawal and statin therapy.

#### **Exclusion Criteria**

Subjects who satisfy any of the following exclusion criteria will be ineligible for enrollment:

- 1. Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to Screening Visit 1 (significant alcohol consumption is defined as more than 2 units/day in females and more than 4 units/day in males, on average).
- 2. Prior intolerance to treatment with atorvastatin or other 3-hydroxy-3-methyl-glutaryl (HMG) Coenzyme A reductase inhibitors (including but not limited to rhabdomyolysis).
- 3. LDL cholesterol ≥190 mg/dL and already on statin therapy at Screening Visit 1.
- 4. LDL cholesterol >200 mg/dL at any Screening visit in subjects who are not on statin therapy, or at Screening Visit 2 in statin washout subjects.
- 5. Planned change in diet or exercise habits during participation in the double-blind period, or a significant weight change of >5% in the prior 6 months.
- 6. Subjects who have undergone gastric bypass procedures (gastric lap band is acceptable) or ileal resection or plan to undergo either of these procedures.
- 7. History of biliary diversion.
- 8. Uncontrolled diabetes defined as  $HbA1c \ge 9.5\%$  within 60 days prior to randomization (Day 1).
- 9. Administration of any of the following medications as specified below:
  - Prohibited <u>30 days</u> prior to Day 1:
    - bile acid sequestrants including cholestyramine and it's derivatives, colesevelam, colestipol, or
    - omega-3 fatty acid-containing dietary supplements
  - Prohibited 3 months prior to Day 1:
    - nicotinic acid and derivatives, ezetimibe, or
    - any prescription or over-the-counter medication or herbal remedy with putative NASH efficacy (except Vitamin E or TZDs), or
    - ursodeoxycholic acid, or
    - fenofibrate or other fibrates, or
    - Any over-the-counter or health foods used to treat lipids including plant sterols and berberine
  - Prohibited 6 months prior to Day 1:
    - azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate, mofetil, pentoxifylline;
       budesonide and other systemic corticosteroids, or
    - potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin)

- Prohibited 12 months prior to Day 1:
  - antibodies or immunotherapy directed against interleukins, or
  - other cytokines or chemokines
- 10. Evidence of other forms of known chronic liver disease including but not limited to:
  - Positive test result at Screening for hepatitis B surface antigen
  - Active hepatitis C virus (HCV) infection (positive for HCV ribonucleic acid [RNA] at Screening) or history of positive HCV RNA test result
  - Primary biliary cirrhosis (also known as primary biliary cholangitis), primary sclerosing cholangitis, autoimmune hepatitis or overlap syndrome
  - Alcoholic liver disease
  - Wilson's disease or hemochromatosis or iron overload as defined by presence of 3+ or 4+ stainable iron on liver biopsy
  - Alpha-1-antitrypsin (A1AT) deficiency as defined by diagnostic features in liver histology (confirmed by A1AT level less than normal; exclusion at the Investigator's discretion)
  - Prior known drug-induced liver injury within 5 years before Day 1
  - Known or suspected hepatocellular carcinoma
- 11. History of liver transplant, current placement on a liver transplant list, or current Model for End-Stage Liver Disease (MELD) score >12. Subjects who are placed on a transplant list despite a relatively early disease stage (eg, per regional guidelines) may be eligible as long as they do not meet any of the other exclusion criteria.
- 12. Presence of hepatic decompensation, including:
  - Gastroesophageal varices
  - Ascites
  - Hepatic encephalopathy
  - Spontaneous bacterial peritonitis
  - Hepatorenal or hepatopulmonary syndromes
- 13. Total bilirubin ≥2x upper limit of normal (ULN) at any Screening visit (subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >2x ULN if their conjugated bilirubin is <2x ULN).
- 14. Creatine phosphokinase >5x ULN at Screening Visit 2.
- 15. Serum creatinine ≥1.5 mg/dL at any Screening visit.
- 16. Serum ALT >300 U/L at any Screening visit.
- 17. Platelet count <75 000/mm3 at any Screening visit.
- 18. Known positivity for human immunodeficiency virus (HIV) infection.
- 19. Subjects with recent history (within 1 year of randomization) of cardiovascular disease or with history or planned cardiovascular interventions to treat atherosclerotic cardiovascular disease, including:
  - a. Peripheral or Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting)
  - b. Coronary angioplasty, stenting, or carotid atherectomy
  - c. Cardiac pacemaker or defibrillator (placement of cardiac pacemaker or defibrillator for reasons other than atherosclerotic cardiovascular disease [eg, for treatment of atrial fibrillation subsequent to nodal ablation] is not exclusionary)

- d. Prosthetic heart valves
- e. Myocardial infarct, unstable angina, or acute coronary syndrome
- f. Other clinically significant atherosclerotic cardiovascular disease
- g. Cerebrovascular accident (stroke), cerebrovascular ischemia, or transient ischemic attack
- h. Unstable hypertension
- i. Familial hypercholesterolemia or other genetic lipid abnormality
- 20. Other concomitant disease, malignancy, or condition likely to significantly decrease life expectancy to <5 years, including known cancers (except carcinomas in situ or other stable, relatively benign conditions such as chronic lymphocytic leukemia) and moderate to severe congestive heart failure.
- 21. Known substance abuse, including inhaled or injected drugs in the year before Screening.
- 22. For female subjects: pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the study, or breastfeeding.
- 23. Participation in a clinical research study with any investigational product being evaluated for the treatment of diabetes or NASH in the 6 months before Day 1.
- 24. Receipt of any investigational product not being evaluated for the treatment of diabetes or NASH from Screening Visit 1 to Day 1, within 30 days prior to Day 1, or within 5 half-lives of the compound before Day 1 (whichever was longer).
- 25. Previous exposure to OCA.
- 26. History of known or suspected clinically significant hypersensitivity to OCA or any of its components.
- 27. Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
- 28. Any other condition which, in the opinion of the Investigator, would impede compliance or hinder completion of the study.
- 29. Acute cholecystitis or acute biliary obstruction

## **Investigational Product, Dosage and Mode of Administration:**

OCA: 5 mg, 10 mg, or 25 mg or placebo tablets, once daily, oral administration

### Study Medication, Dosage and Mode of Administration:

Atorvastatin: 10 mg, 20 mg, 40 mg, 80 mg once daily, oral administration

#### **Duration of Subject Participation:**

- Screening period for statin-using subjects: Up to 5 weeks (including a 4-week statin washout period)
- Screening period for non-statin-using subjects: Up to 5 weeks
- Double-Blind period: 16 weeks

• LTSE: 2 years

#### **Duration of Treatment:**

#### **Double-Blind period**:

OCA/placebo: 16 weeks (Day 1 to Week 16)

Atorvastatin: 12 weeks (Week 4 to Week 16), administered open-label

### LTSE:

OCA: 2 years

• Atorvastatin: As clinically indicated

#### Reference Therapy, Dosage and Mode of Administration:

Not applicable

#### **Criteria for Evaluation:**

#### **Statistical Methods:**

The assessments supporting the primary, secondary, and exploratory objectives of the study are as follows:

| Primary Endpoints | Assessment |
|---|---|
| LDL metabolism | LDL cholesterol concentration, particle size, and particle concentration |
| Secondary Endpoints | |
| Lipoprotein metabolism | HDL cholesterol concentration, particle size and particle concentration; VLDL cholesterol concentration, particle size and particle concentration; TG and total cholesterol concentrations; apolipoprotein (Apo)A1, ApoB, ApoE, ApoCII, ApoCIII and Lp(a) concentrations; PCSK9 concentration |
| Reverse cholesterol transport | Pre-β1 HDL concentration, macrophage cholesterol efflux; LCAT activity; CETP activity |
| Safety and tolerability | TEAEs (including cardiovascular events), physical exams, ECGs, vital signs, clinical laboratory assessments (including lipid profile changes) |
| <b>Exploratory Endpoints</b> | |
| Liver biochemistry and markers of liver function | Albumin, ALP (isoenzymes), ALT, AST, , direct bilirubin, GGT, INR, total bilirubin |
| Markers of liver inflammation | IL-6, hs-CRP, and TNF-α |
| Marker for hepatic apoptosis and fibrosis | CK-18-M30 and CK-18-M65 |
| Glycemic Control | Glucose, insulin, C-peptide, HbA1c, HOMA-β, and HOMA-IR |
| OCA pharmacokinetics | OCA, tauro-OCA, glyco-OCA, total OCA, potentially other conjugates or metabolites not yet identified |
| Atorvastatin bioanalytical concentrations | Atorvastatin and its metabolites |
| Anthropometric measures | Height (at Screening Visit 1 only), weight, and waist and hip circumference measurements; and body mass index (BMI), and waist-to-hip ratio calculations |
| Pharmacodynamics | C4 (7α-hydroxy-4-cholesten-3-one), and FGF-19; possible analysis of conjugated and unconjugated endogenous bile acids |
| Noninvasive radiological liver fibrosis measurements | By TE (where available) |
| Cardiovascular risk scores | FRS and Reynolds scores |

ALP = alkaline phosphatase; ALT = alanine aminotransferase; ApoA1 = apolipoprotein A1; ApoB = apolipoprotein B; ApoCII = apolipoprotein CII; ApoCIII = apolipoprotein CIII; ApoE = apolipoprotein E; AST = aspartate aminotransferase; BMI = body mass index; C4 =  $7\alpha$ -hydroxy-4-cholesten-3-one; CK-18-M30 = cytokeratin-18 neoepitope M30; CK-18-M65 = cytokeratin-18 neoepitope M65; CTEP = cholesterol ester transfer protein; FGF-19 = fibroblast growth factor-19; FRS = Framingham Risk Score; GGT = gamma-glutamyl transferase; HbA1c = hemoglobin-specific A1c fraction; HDL = high-density lipoprotein; HOMA- $\beta$ : homeostatic model assessment – beta-cell function; HOMA-IR = homeostatic model assessment – insulin resistance; hs-CRP = high sensitivity C-reactive protein; IL-6 = interleukin-6; INR = international normalized ratio; LCAT = lecithin cholesterol acyltransferase; LDL = low-density lipoprotein; Lp(a) = lipoprotein(a); PCSK9 = proprotein convertase subtilisin/kexin type 9; PD = pharmacodynamics; TE = transient elastography; TEAE = treatment emergent adverse event; TG = triglyceride; TNF- $\alpha$  = tumor necrosis factor- $\alpha$ ; VLDL = very low-density lipoprotein

#### **Analysis Populations:**

The following analysis populations will be used:

## Intent-to-Treat (ITT) Population

All randomized subjects who receive any amount of investigational product will be included in the ITT Population. Treatment assignment will be based on the randomized treatment allocation.

#### Safety Population

The Safety Population will include all subjects who receive any amount of investigational product. Treatment assignment will be based on the treatment actually received. The Safety Population will be used for the analysis of all safety data.

## **Efficacy Evaluable Population**

All subjects who complete the double-blind phase according to the indicated doses of investigational product and atorvastatin without any significant protocol deviations. The Efficacy Evaluable Population will be the primary population used for efficacy analyses.

#### Pharmacokinetic Populations

The OCA PK Population will include all OCA subjects who consent to participate in the PK assessments and have at least one confirmed fasted analyzable sample. Subjects must have been fasting for approximately 8 hours before the visit and must not have any major protocol deviations that potentially affect exposure levels. The Atorvastatin PK Population will include all subjects who consent to participate in the PK assessments and have at least one confirmed fasted analyzable sample.

#### LTSE Population

All subjects who receive any amount of investigational product as part of the LTSE will be included in the LTSE Population.

#### **Efficacy Analyses:**

The primary efficacy analyses will be based on the Efficacy Evaluable Population.

The primary efficacy parameter, changes in LDL cholesterol, particle size and particle concentration at Week 16 (end of the double-blind phase) compared to Baseline will be summarized by treatment group.

Analyses of observed LDL values will be carried out using an analysis of covariance (ANCOVA) model at each visit with change from baseline as the dependent variable, including treatment group and randomization stratification factor as fixed effects and baseline as a covariate. The same analysis will be carried out using percentage change from baseline as the dependent variable.

Descriptive statistics of the values will be summarized by treatment group and visit. The results, change from baseline, and percentage change from baseline values as well as estimates of least-square (LS) means, standard errors, and 95% confidence intervals (CIs) will be presented by treatment group.

The comparison of LDL change from baseline and percentage change from baseline values between each active treatment group and placebo group will be performed as exploratory analysis. Estimates of the LS mean difference between each active treatment group and placebo group, the standard error of the difference, and 95% CI of the difference will be presented.

The secondary parameters will be analyzed in the same manner as the primary efficacy variables. Descriptive statistics will be generated and will include change from baseline, percentage change from baseline, and estimates of LS means, standard errors, and 95% CIs presented by treatment group.

The secondary parameters related to lipoprotein metabolism include HDL cholesterol concentration, particle size and particle concentration; VLDL cholesterol concentration, particle size and particle concentration; TG and total cholesterol concentrations; and apolipoprotein (Apo)A1, ApoB, ApoE, ApoCII, ApoCIII and Lp(a) concentrations.

The secondary parameters related to reverse cholesterol metabolism include pre-β1 HDL concentration, macrophage cholesterol efflux; lecithin cholesterol acyltransferase (LCAT) activity; and cholesterol ester transfer protein (CETP) activity.

The baseline value for efficacy analyses is defined as the last value prior to administration of investigational product on Day 1 (predose).

The following exploratory parameters will be analyzed in the same manner as the secondary efficacy variable: markers of liver biochemistry, liver function, liver inflammation, apoptosis, liver fibrosis, glycemic control, and bile acids. Additionally, descriptive statistics will be generated and will include change from baseline, percentage change from baseline, and estimates of LS means, standard errors, and 95% CIs presented by treatment group. Changes from baseline will be summarized for anthropometric measures. PK analysis will be done using non-compartmental methods. The values will be summarized by active treatment group using descriptive statistics. Only samples that have a confirmed fasting of approximately 8 hours or more before their visit will be included in the PK analysis. Further details regarding specific parameters and methods will be described in the Statistical Analysis Plan.

#### **Safety Analyses:**

All safety analyses will be based on the Safety Population. The incidence of treatment-emergent adverse events (TEAEs) and serious AEs (SAEs) will be tabulated by system organ class and preferred term for each treatment group, and similarly by severity and relationship to treatment. The incidence of pre-treatment AEs and pre-treatment SAEs occurring after informed consent form signoff and before the first dosing of investigational product (OCA or placebo) will be tabulated in the same manner as above for all subjects participating in the washout period.

Laboratory parameters, physical examinations including vital signs, and ECGs will be summarized by treatment group using descriptive statistics at Baseline and at each scheduled post-Baseline visit. The absolute change from baseline will also be summarized.

#### LTSE Analyses:

Similar analyses to that which are described above will be conducted for the LTSE using the double-blind baseline value. Analyses based on the double-blind baseline will be performed using randomized treatment groups (placebo, OCA 5 mg, OCA 10 mg, or OCA 25 mg). Sensitivity analyses may be conducted using the last value prior to first dose in the LTSE for all subjects.

#### **Sample Size Justification:**

It is the intent of this study to characterize the components of LDL metabolism (cholesterol concentration, particle size, particle concentration) in subjects with NASH before and after treatment with OCA and to assess the changes induced by HMG Coenzyme A reductase inhibitor (atorvastatin) therapy. Assuming a 22 mg/dL increase from baseline with a standard deviation of 24 in LDL in the OCA 25 mg group without atorvastatin therapy after 16 weeks of treatment based on data from FLINT, a sample size of 20 subjects per group will provide greater than 97.3% power to demonstrate the statistically significant difference of LDL increase from baseline with a 2-sided type I error of 0.05.

# 3. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

# **TABLE OF CONTENTS**

| 1. | TITLE PAGE | |
|---|---|---|
| 2. | SYNOPSIS | |
| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 14 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 22 |
| 5. | INTRODUCTION | 26 |
| 5.1. | Overview of Nonalcoholic Steatohepatitis and Obeticholic Acid | 26 |
| 5.2. | NASH, Lipoprotein Metabolism, and Statins | 27 |
| 5.3. | Mechanism of Action of Obeticholic Acid | 28 |
| 5.4. | Nonclinical Experience with Obeticholic Acid | 29 |
| 5.5. | Clinical Experience with Obeticholic Acid | 30 |
| 5.6. | Rationale for Study Design, Doses of Investigational Product and Use of Atorvastatin. | 32 |
| 5.6.1. | Rational for Study Design | 32 |
| 5.6.2. | Rationale for Placebo Control Group | 33 |
| 5.6.3. | Rationale for OCA Doses | 33 |
| 5.6.4. | Rationale for the Use of Atorvastatin | 34 |
| 5.6.4.1. | Rationale for Statin Withdrawal | 34 |
| 5.6.5. | Rationale for Duration of Treatment | 35 |
| 5.6.6. | Rationale for Timing of Unblinding Process and Implications in LTSE | 36 |
| 5.7. | Summary of Known Potential Risks with Investigational Product | 36 |
| 5.8. | Summary of Known Potential Risks with Atorvastatin | 36 |
| 6. | STUDY OBJECTIVES AND PURPOSE | 38 |
| 6.1. | Primary Objective | 38 |
| 6.2. | Secondary Objectives | 38 |
| 6.3. | Exploratory Objectives | 38 |
| 7. | INVESTIGATIONAL PLAN | 39 |
| 7.1. | Overall Study Design | 39 |
| 7.1.1. | Study Design | 40 |
| 7.1.2. | Schedule of Study Procedures | 41 |
| 7.1.3. | Study Duration | 46 |

| 7.2. | Number of Subjects | 46 |
|---|---|---|
| 7.3. | Treatment Assignment | 46 |
| 7.4. | Dose Adjustment Criteria | 46 |
| 7.4.1. | Investigational Product Dose Adjustments | 46 |
| 7.4.2. | Atorvastatin Dose Adjustments | 46 |
| 7.4.3. | Safety Criteria for Adjustment or Stopping of Doses of Investigational Product | 47 |
| 7.5. | Criteria for Study Termination | 48 |
| 8. | SELECTION AND WITHDRAWAL OF SUBJECTS | 48 |
| 8.1. | Subject Population | 48 |
| 8.2. | Subject Inclusion Criteria | 48 |
| 8.3. | Subject Exclusion Criteria | 49 |
| 8.4. | Subject Withdrawal Criteria | 52 |
| 8.4.1. | Reasons for Mandatory Discontinuation of Investigational Product or Atorvastatin. | |
| 8.4.1.1. | Adverse Events \(\geq\)Grade 3 in Severity and Possibly, Probably, or Definitely Related to Investigational Product. | 52 |
| 8.4.1.2. | Pregnancy | 52 |
| 8.4.1.3. | Severe Drug-Induced Liver Injury | 52 |
| 8.4.1.4. | Myonecrosis | 53 |
| 8.4.2. | Reasons for Mandatory Interruption of Investigational Product | 53 |
| 8.4.2.1. | Adverse Events \(\geq\)Grade 4 in Severity and Not or Unlikely Related to Investigational Product | 53 |
| 8.4.2.2. | Suspected Mild or Moderate Drug-Induced Liver Injury | 53 |
| 8.4.3. | Other Reasons for Study or Treatment Discontinuation of Subjects | 54 |
| 8.4.4. | Subject Discontinuation Notification | 54 |
| 9. | TREATMENT OF SUBJECTS | 54 |
| 9.1. | Investigational Product and Atorvastatin Treatment Regimen | 54 |
| 9.1.1. | Double-Blind Period | 55 |
| 9.1.2. | LTSE | 55 |
| 9.2. | Concomitant Medications | 55 |
| 9.2.1. | Medications with Potential NASH-Modifying Properties | 55 |
| 9.2.2. | Diabetes-Specific Therapy | 56 |
| 9.2.3. | Management of Changes in Cholesterol | 56 |

| - | | Page 1 |
|---|---|---|
| 9.2.4. | Prohibited Medications | 56 |
| 9.2.5. | Standard of Care and Other Concomitant Medications | 60 |
| 9.3. | Treatment Compliance | 60 |
| 9.4. | Randomization and Blinding | 60 |
| 9.4.1. | Stratification | 61 |
| 9.4.2. | Emergency Unblinding Procedures | 61 |
| 9.5. | Assignment of Site and Subject Numbers | 62 |
| 9.5.1. | Site Numbers | 62 |
| 9.5.2. | Subject Numbers | 62 |
| 9.6. | Restrictions | 62 |
| 9.6.1. | Fasting Requirement at Study Visits | 62 |
| 9.6.2. | Grapefruit and Grapefruit Juice | 62 |
| 9.6.3. | Diet and Exercise | 62 |
| 9.7. | Visit Procedures | 62 |
| 9.7.1. | | |
| 9.7.2. | 7.2. Informed Consent Procedures. | |
| 9.7.3. | Screening Visit 1 Procedures | 64 |
| 9.7.4. | Screening Visit 2 Visit Procedures | 65 |
| 9.7.5. | Randomization/Day 1 Visit Procedures | 65 |
| 9.7.6. | Week 2 Visit Procedures | 67 |
| 9.7.7. | Week 4 Visit Procedures | 68 |
| 9.7.8. | Week 6 Safety Contact | 69 |
| 9.7.9. | Week 8 Visit Procedures | 69 |
| 9.7.10. | Week 10 Safety Contact | 70 |
| 9.7.11. | Week 12 Visit Procedures | 71 |
| 9.7.12. | Week 14 Safety Contact | 72 |
| 9.7.13. | Week 16 Visit Procedures | 72 |
| 9.7.13.1. | Additional Week 16 Procedures for PK Subjects | 73 |
| 9.7.14. | Additional Procedures at Week 16/LTSE Day 1 Visit for Subjects Continuing into the LTSE | 73 |
| 9.7.15. | Early Termination/End of Study Procedures: Double-Blind Period | |
| 9.7.16. | LTSE Visits | |

9.7.17.

| 9.7.18. | LTSE Month 3, Month 6, Month 9, Month 15, Month 18, and Month 21 Visit Procedures | 77 |
|---|---|---|
| 9.7.19. | LTSE Month 12 Visit Procedures | 78 |
| 9.7.20. | LTSE End of Study/Early Termination Procedures | 79 |
| 9.7.21. | Unscheduled Safety Visits | 81 |
| 10. | INVESTIGATIONAL PRODUCT AND STUDY MEDICATION | 81 |
| 10.1. | Investigational Product (OCA or Placebo) | 81 |
| 10.2. | Investigational Product Packaging and Labeling | 81 |
| 10.3. | Investigational Product Storage | 82 |
| 10.4. | Investigational Product Administration | 82 |
| 10.4.1. | Investigational Product Dispensation | 82 |
| 10.4.2. | Missed Doses | 82 |
| 10.5. | Atorvastatin Tablets | 82 |
| 10.5.1. | Atorvastatin Packaging and Labeling | 83 |
| 10.5.1.1. | Atorvastatin Storage | 83 |
| 10.5.2. | Atorvastatin Administration | 83 |
| 10.5.3. | Atorvastatin Dispensation | |
| 10.5.4. | Missed Doses of Atorvastatin | 83 |
| 10.5.5. | Atorvastatin Overdose | 83 |
| 10.6. | Investigational Product and Atorvastatin Accountability and Disposal | 84 |
| 11. | ASSESSMENT OF EFFICACY AND PHARMACOKINETICS | 84 |
| 11.1. | Efficacy Assessments | 84 |
| 11.1.1. | Efficacy Laboratory Assessments | 86 |
| 11.1.2. | Liver Biopsy | 86 |
| 11.1.2.1. | Central Reading of Liver Histology | 86 |
| 11.1.3. | Noninvasive Radiological Liver Fibrosis Measurements | 87 |
| 11.1.4. | Blood Samples for Future Analysis | 87 |
| 11.2. | Pharmacokinetic and Pharmacodynamic Assessments | 87 |
| 11.2.1. | Pharmacodynamic Assessments | 87 |
| 11.2.2. | Pharmacokinetic Assessments | 88 |
| 11.3. | Anthropometric Assessments | 88 |
| 11.3.1. | BMI | 88 |
| 11.3.2. | Body Weight | 88 |

| 11.3.3. | Waist and Hip Circumference: | 88 |
|---|---|---|
| 12. | ASSESSMENT OF SAFETY | 89 |
| 12.1. | Adverse Events and Serious Adverse Events | 89 |
| 12.1.1. | Definitions | 89 |
| 12.1.1.1. | Adverse Event | 89 |
| 12.1.1.2. | Treatment-Emergent Adverse Event | 89 |
| 12.1.1.3. | Serious Adverse Event | 89 |
| 12.1.2. | Relationship to Investigational Product or Study Medication | 90 |
| 12.1.3. | Relationship to Liver Biopsy | 91 |
| 12.1.4. | Recording Adverse Event Severity | 91 |
| 12.1.4.1. | Severity of Pruritus (as an AE) | 92 |
| 12.1.5. | Reporting of Adverse Events and Serious Adverse Events | 93 |
| 12.1.5.1. | Reporting of Adverse Events | 93 |
| 12.1.5.2. | Reporting of Serious Adverse Events | 93 |
| 12.1.6. | Additional Investigator Responsibilities for SAEs | 94 |
| 12.1.7. | Notification of Post-Study SAEs | 94 |
| 12.1.8. | Follow-Up of Adverse Events and Serious Adverse Events | 95 |
| 12.1.8.1. | Pregnancy and Follow-Up | 95 |
| 12.2. | Other Safety Parameters | 96 |
| 12.2.1. | Medical History/Demographics | 96 |
| 12.2.2. | Physical Examination | 96 |
| 12.2.3. | Vital Signs | 96 |
| 12.2.4. | Electrocardiogram | 96 |
| 12.2.5. | Alcohol Consumption | 97 |
| 12.2.6. | Laboratory Assessments | 97 |
| 13. | STATISTICS | 99 |
| 13.1. | Analysis Sets | 99 |
| 13.2. | Determination of Sample Size | 100 |
| 13.3. | General Statistical Considerations | 100 |
| 13.4. | Handling of Dropout and Missing Data | 100 |
| 13.5. | Subject Population and Demographic Characteristics | 100 |
| 13.6. | Efficacy Analysis | 100 |

| 13.6.1. | Primary Efficacy Analysis | 101 |
|---|---|---|
| 13.6.2. | Secondary Efficacy Analysis | 101 |
| 13.6.3. | Additional Exploratory Efficacy Analyses | 101 |
| 13.6.3.1. | Liver Biochemistry, Hepatobiliary Damage, and Liver Function | 101 |
| 13.6.3.2. | Markers of Inflammation, Fibrosis, and/or Apoptosis | 102 |
| 13.6.3.3. | Glycemic Control Measures | 102 |
| 13.6.3.4. | Anthropometric Measures and Blood Pressure | 102 |
| 13.6.3.5. | Noninvasive Radiological Liver Fibrosis Measurements | 103 |
| 13.6.3.6. | Pharmacodynamic Analysis. | 103 |
| 13.6.3.7. | Pharmacokinetic Analysis | 103 |
| 13.6.3.8. | Cardiovascular Risk Scores | 103 |
| 13.6.4. | LTSE Analyses | 104 |
| 13.7. | Safety Analysis | 104 |
| 13.7.1. | Adverse Events | 104 |
| 13.7.2. | Clinical Laboratory Evaluations | 104 |
| 13.7.3. | Lipoprotein Evaluations | 104 |
| 13.7.4. | Additional Safety Analysis | 105 |
| 13.7.4.1. | Vital Signs | 105 |
| 13.7.4.2. | Electrocardiograms | 105 |
| 13.7.5. | Adjudicated Cardiovascular Events | 105 |
| 13.8. | Data Monitoring Committee | 105 |
| 13.9. | Adjudication Committees | 106 |
| 14. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 107 |
| 14.1. | Study Monitoring | 107 |
| 14.2. | Audits and Inspections | 107 |
| 15. | QUALITY CONTROL AND QUALITY ASSURANCE | 107 |
| 16. | ETHICS | 108 |
| 16.1. | Ethics Review | 108 |
| 16.2. | Ethical Conduct of the Study | 108 |
| 16.3. | Written Informed Consent | 108 |
| 16.4. | Subject Confidentiality and Data Protection | 109 |
| 17 | INVESTIGATOR OBLIGATIONS | 109 |

| 17.1. | AE Reporting1 | |
|---|---|---|
| 17.2. | Protocol Deviations | |
| 17.3. | Regulatory Documentation | |
| 17.4. | Ethics Review | 110 |
| 17.5. | Archiving and Record Retention | 110 |
| 18. | PUBLICATION POLICY | 111 |
| 19. | LIST OF REFERENCES. | 113 |
| APPENDI | X A. AMERICAN COLLEGE OF CARDIOLOGY/AMERICAN HEART ASSOCIATION GUIDANCE FOR THE USE OF STATINS | 118 |
| APPENDI | X B. GUIDANCE FOR ELEVATED LIVER BIOCHEMISTRY VALUES | 165 |
| APPENDI | X C. COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS | 167 |
| APPENDI | X D. STANDARDIZED DEFINITIONS FOR CARDIOVASCULAR ENDPOINT EVENTS | 248 |
| APPENDI | X E. ATORVASTATIN PRESCRIBING INFORMATION | 277 |
| APPENDI | X F. 747-209 PROTOCOL VERSION 2 SUMMARY OF CHANGES | 310 |
| APPENDI | X G. 747-209 PROTOCOL VERSION 3 SUMMARY OF CHANGES | 335 |
| APPENDI | X H. 747-209 PROTOCOL VERSION 4 SUMMARY OF CHANGES | 359 |
| | LIST OF TABLES | |
| Table 1: | Schedule of Study Procedures: Double-Blind Period | 41 |
| Table 2: | Schedule of Study Procedures: LTSE | 44 |
| Table 3: Medications Prohibited Prior to Randomization and/or During Study Participation | | 58 |
| Table 4: | • | |
| Table 5: | Table 5: NASH CRN Scoring System for Determining Eligibility and Primary Histological Endpoint Assessment | |
| Table 6: | Table 6: Relationship of Adverse Events to Investigational Product or Study Medication | |
| Table 7: | Relationship of Adverse Events to Liver Biopsy | 91 |
| Table 8: | Severity of Adverse Events | 92 |
| Table 9: | Severity of Pruritus | 92 |
| Table 10: | List of Laboratory Analytes to be Tested | |

# LIST OF FIGURES

| Figure 1: | Study Design Schematic | 40 |
|-----------|------------------------|----|
| 8 | ~ ****** | |

# 4. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this protocol.

| Abbreviation or Specialist Term | Explanation |
|---|---|
| 6-ECDCA | 6α-ethyl-chenodeoxycholic acid |
| A1AT | alpha-1-antitrypsin |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| ApoA1 | apolipoprotein A1 |
| ApoB | apolipoprotein B |
| ApoCII | apolipoprotein CII |
| ApoCIII | apolipoprotein CIII |
| АроЕ | apolipoprotein E |
| AST | aspartate aminotransferase |
| β-hCG | beta human chorionic gonadotropin |
| BAS | bile acid sequestrants |
| BMI | body mass index |
| BNP | B-type natriuretic peptide |
| BUN | blood urea nitrogen |
| C4 | 7α-hydroxy-4-cholesten-3-one |
| CAC | Cardiovascular Adjudication Committee |
| CDCA | chenodeoxycholic acid |
| CETP | cholesterol ester transfer protein |
| CI | confidence interval |
| CK-18-M30 | cytokeratin-18 neoepitope M30 |
| CK-18-M65 | cytokeratin-18 neoepitope M65 |
| COX-2 | cyclooxygenase-2 |
| СРК | creatine phosphokinase |
| CRA | Clinical Research Associate |
| CRF | case report form(s) |
| CRN | clinical research network |
| CTCAE | Common Terminology Criteria for Adverse Events |

| Abbreviation or Specialist Term | Explanation |
|---|---|
| DMC | Data Monitoring Committee |
| eCRF | electronic case report form(s) |
| ECG | electrocardiogram |
| EDC | electronic data capture |
| EOS | End of Study |
| ET | Early Termination |
| FGF-19 | fibroblast growth factor-19 |
| FLINT | Farnesoid X Receptor Ligand Obeticholic Acid in NASH<br>Treatment |
| FRS | Framingham Risk Score |
| FXR | farnesoid X receptor |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| glyco-OCA | glycine conjugate of OCA |
| GMP | Good Manufacturing Practice |
| HbA1c | hemoglobin-specific A1c fraction |
| HCC | hepatocellular carcinoma |
| HDL | high-density lipoprotein |
| HDLc | high-density lipoprotein cholesterol |
| HDPE | High-density polyethylene |
| HIV | human immunodeficiency virus |
| HMG | 3-hydroxy-3-methyl-glutaryl |
| НОМА-β | homeostatic model assessment-beta-cell function |
| HOMA-IR | homeostatic model assessment – insulin resistance |
| hs-CRP | high-sensitivity C-reactive protein |
| IB | Investigator's Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| IEC | Independent Ethics Committee |
| IND | investigational new drug |
| iNOS | inducible nitric oxide synthase |

| Abbreviation or Specialist Term | Explanation |
|---|---|
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| ISF | Investigator site file |
| ITT | intent-to-treat |
| IWRS | interactive web response system |
| LCAT | lecithin cholesterol acyltransferase |
| LDL | low-density lipoprotein |
| LDLc | low-density lipoprotein cholesterol |
| Lp(a) | lipoprotein(a) |
| LS | least-square |
| LTSE | long-term safety extension |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MELD | Model for End-Stage Liver Disease |
| NAFLD | nonalcoholic fatty liver disease |
| NAS | nonalcoholic fatty liver disease activity score |
| NASH | nonalcoholic steatohepatitis |
| NMR | nuclear magnetic resonance |
| OCA | obeticholic acid |
| PAI-1 | plasminogen activator inhibitor-1 |
| PBC | primary biliary cirrhosis (also known as primary biliary cholangitis |
| PCSK9 | proprotein convertase subtilisin/kexin type 9 |
| PD | pharmacodynamics(s) |
| PI | Principal Investigator |
| PK | pharmacokinetic(s) |
| PSC | primary sclerosing cholangitis |
| QTcF | QT interval corrected by Fridericia's formula |
| SAE | serious adverse event |
| SAP | Statistical Analysis Plan |
| SAR | suspected adverse reaction |
| SREBP1c | sterol regulatory element binding protein |
| SUSAR | suspected unexpected serious adverse reaction |

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|----------------------------------|
| Т3 | triiodothyronine |
| T4 | thyroxine |
| tauro-OCA | taurine conjugate of OCA |
| TE | transient elastography |
| TEAE | treatment-emergent adverse event |
| TG | triglyceride |
| TNF-α | tumor necrosis factor-α |
| TSH | thyroid-stimulating hormone |
| ULN | upper limit of normal |
| VLDL | very low-density lipoprotein |

#### 5. INTRODUCTION

# 5.1. Overview of Nonalcoholic Steatohepatitis and Obeticholic Acid

Nonalcoholic fatty liver disease (NAFLD) is considered to be the hepatic manifestation of metabolic syndrome, a cluster of closely related clinical features linked to visceral obesity and characterized by insulin resistance, dyslipidemia, and hypertension (Chalasani 2012, Angulo 2011). NAFLD is the most common cause of chronic liver disease in the western hemisphere, and as the prevalence of obesity and metabolic syndrome rises, a parallel rise of NAFLD across the world is generally expected. NAFLD is thought to be represented by a spectrum of histological disease, which progresses from pure fatty liver (simple steatosis) to nonalcoholic steatohepatitis (NASH). While NAFLD itself is considered a relatively benign and reversible condition, up to one-third of patients in the spectrum of NAFLD develop NASH, a chronic, serious, life-threatening, inflammatory liver disease characterized by hepatocellular injury, inflammation, and progressive fibrosis. As opposed to simple steatosis, NASH is associated with significant morbidity and progression that, if left untreated, can progress to advanced fibrosis, cirrhosis, hepatic decompensation, hepatocellular carcinoma (HCC), and liver-related death (Vernon 2011).

Of all the histologic features of NASH, fibrosis is considered the strongest predictor of adverse clinical outcomes, including liver-related death (Younossi 2011, Ekstedt 2014). Patients with NASH develop progressive fibrosis over a period of 4 to 6 years (Pagadala 2012) and 21% to 26% of these patients develop cirrhosis in 8.2 years (Loomba 2013). In patients with NASH who have progressed to cirrhosis, it is estimated 38% to 45% have liver failure after 7 years to 10 years, and 2% to 5% of this population will develop HCC per year (Organisation 2012). Accumulating evidence suggests that patients with NASH can progress to HCC, even in the absence of apparent cirrhosis (Williams 2013, Ertle 2011).

There are currently no approved therapies for the treatment of NASH nor an accepted standard of care. The therapeutic options for NASH are largely limited to lifestyle modifications and treatment of concurrent conditions such as diabetes (Chalasani 2012, Neuschwander-Tetri 2003, Sanyal 2010, Belfort 2006), although practice guidelines from the American Association for the Study of Liver Diseases recommend the use of vitamin E as first line therapy for patients with NASH without diabetes.

In view of the serious nature of the disease, the increasing prevalence, the complications that arise from the disease, and the clear unmet medical need, evaluation of therapies for NASH is warranted.

Obeticholic acid (OCA) is a modified bile acid and farnesoid X receptor (FXR) agonist that is derived from the primary bile acid chenodeoxycholic acid (CDCA). CDCA is the natural ligand for FXR, which is a nuclear receptor expressed at high levels in the liver, intestine, kidney, and adrenal glands. In the liver, FXR is expressed in hepatocytes, Kupffer cells, and endothelial cells, and at a low level in hepatic stellate cells. Nuclear receptors constitute a family of ligand-activated transcription factors that can either activate or repress a variety of target genes.

OCA is 100-fold more potent than the endogenous FXR agonist CDCA, which makes OCA an attractive novel therapeutic agent for NAFLD and NASH due to its multiple FXR-mediated effects, including an increase in insulin sensitivity, glucose and lipid metabolism; hepatocyte

protection against bile acid-induced cytotoxicity; anti-inflammatory effects in liver and vasculature; and prevention and reversal of liver fibrosis (Mudaliar 2013, Adorini 2012). Thus, there is strong rationale to advance OCA for the treatment of NASH based on its FXR-mediated hepatoprotective properties, and results that indicate OCA improves glycemia by increasing peripheral glucose uptake, enhances glucose-stimulated insulin secretion, and inhibits hepatic lipid synthesis and content while inducing lipid uptake by adipocytes.

# 5.2. NASH, Lipoprotein Metabolism, and Statins

NAFLD is the most common cause of incidental abnormal serum liver enzymes and is associated with dyslipidemia and high-risk of cardiovascular events. Statins have been shown to reduce the risk of major coronary and vascular events in NAFLD (Pastori 2015). There has been some concern that patients with underlying liver disease are at an increased risk of hepatotoxicity because the statins are hepatically cleared and can cause elevations in liver enzymes. However, there have also been studies that have shown that elevated serum transaminases secondary to comorbid conditions like NAFLD or NASH may be improved by statin treatment (Athyros 2010, Pastori 2015). Atherogenic hyperlipidemia, which is defined by increased triglycerides (TGs), decreased high-density lipoprotein (HDL), and the presence of small, dense low-density lipoprotein (LDL), is frequently associated with NAFLD, thus the treatment of dyslipidemia plays a critical role in the overall management of NAFLD and NASH.

In the Farnesoid X Receptor Ligand Obeticholic Acid in NASH Treatment (FLINT) Trial conducted by the NASH Clinical Research Network (CRN) at the National Institute of Diabetes and Digestive and Kidney Diseases, subjects with non-cirrhotic NASH were randomized to either placebo or 25-mg OCA for 72 weeks (Neuschwander-Tetri 2014). Subjects in this study were representative of the NASH population with baseline total cholesterol and LDL cholesterol (LDLc) levels at the high end of normal, HDLc levels within the normal range, and TG levels borderline high. Approximately 50% of subjects were receiving antilipidemic agents at Baseline. Increases in total cholesterol, LDLc, and TG were observed in both treatment groups with OCA-treatment being associated with a somewhat greater percentage of subjects exhibiting increased concentrations of total cholesterol and LDLc. Similarly, decreases in HDL cholesterol (HDLc) were observed in both treatment groups with a higher percentage of OCA-treated subjects compared with placebo. While the OCA-related changes in lipids was modest and initial increases in total cholesterol and LDLc trended back towards baseline values with continued treatment, it is important to characterize the mechanism of OCA treatment on lipids in patients with NASH and the functionality of concomitant lipid therapies.

Using nuclear magnetic resonance (NMR) lipid profiling, it will be possible to characterize the effect of OCA on the actual concentration and sizes of the particles within each lipoprotein class. While a standard lipid panel measures the cholesterol or TG content of lipoproteins, it does not measure the actual particle concentration. The cholesterol and TG content of LDL, HDL, and very low-density lipoprotein (VLDL) particles is not constant, but varies widely among individuals and over time. Even within a given lipoprotein class, the sizes of the particles are not uniform as the relative amounts of cholesterol and TG carried in the core of a lipoprotein particle varies across individuals. Compositional differences also relate to plasma TG levels with LDL and HDL particles becoming more cholesterol-depleted and TG-rich as plasma TG levels increase. Thus, presentation of the same measured concentration of LDL in 2 patients may

represent significantly different numbers of LDL particles and, therefore, a different risk for cardiovascular disease (Jeyarajah 2006, Otvos 2006). The patient with the higher number of small, atherogenic LDL particles would be considered to be at higher cardiovascular risk. Thus, NMR lipid profiling, which allows differentiation of particle size and number, will provide a better understanding of the mechanistic impact of OCA treatment on lipids.

Recent evidence also suggests that HDL-mediated atheroprotection is largely governed through regulation of reverse cholesterol transport from macrophages within atherosclerotic plaques to HDL acceptor particles for ultimate return to the liver and biliary excretion (Rohatgi 2014). Thus, this study will also assess macrophage efflux and candidate components of this pathway to further elucidate the mechanism of OCA and atorvastatin treatment on lipids in the presence of NASH.

## 5.3. Mechanism of Action of Obeticholic Acid

CDCA is the principal natural ligand of FXR in humans. When cellular levels are high, the negative feedback pathway inhibits the further synthesis of bile. OCA is structurally related to CDCA and differs by the addition of a single ethyl group (the chemical name of OCA is  $3\alpha 7\alpha$ -dihydroxy- $6\alpha$ -ethyl- $5\beta$ cholan-24-oic acid. It is also referred to as  $6\alpha$ -ethyl-chenodeoxycholic acid, or (6-ECDCA) and as an agonist it is approximately 100-fold more potent than CDCA in vitro (Pellicciari 2002). OCA is also highly selective for FXR and does not bind other nuclear receptors, and with the exception of weakly activating the dedicated bile acid receptor TGR5, it does not activate any G-protein coupled receptors (CEREP 2008).

OCA is an attractive novel therapeutic agent for NAFLD and NASH due to its multiple FXR-mediated effects including an increase in insulin sensitivity, hepatocyte protection against bile acid-induced cytotoxicity, anti-inflammatory effects in liver and vasculature, and prevention and reversal of liver fibrosis (Adorini 2012, Mudaliar 2013). Specifically:

- FXR and other identified bile acid receptors, such as TGR5, play a role in regulating key aspects of carbohydrate and lipid metabolism; thus, serving as important mediators of energy expenditure and metabolic homeostasis.
- FXR agonists have been shown to suppress hepatic fatty acid and TG synthesis through down-regulation of sterol regulatory element binding protein (SREBP1c) and increase hepatic fatty acid oxidation through up-regulation of pyruvate dehydrogenase kinase 4 (Lefebvre 2009).
- FXR activation has insulin-sensitizing effects. In mice fed a high-fat diet, treatment with recombinant fibroblast growth factor-19 (FGF-19) improves indices of dyslipidemia, hepatic steatosis, hyperinsulinemia, hyperleptinemia, and insulin sensitivity, while reducing body weight and adiposity (Fu 2004). Studies in FXR knockout mice show that FXR is involved in the regulation of insulin signaling pathways and the receptor appears to have a beneficial role in decreasing insulin resistance (both hepatic and in skeletal muscle) and gluconeogenesis, as well as in regulating TG, free fatty acid, and lipid levels.

• Treatment of OCA at doses of 25 mg and 50 mg for 6 weeks resulted in increased insulin sensitivity and reduced markers of liver inflammation and fibrosis in subjects with NAFLD and type 2 diabetes mellitus (Mudaliar 2013).

 Treatment with OCA at a dose of 25 mg for 72 weeks was superior to placebo in improving not only the key histologic features important in the underlying pathophysiology of the disease (inflammation, ballooning, steatosis), but notably that OCA was superior to placebo in improving fibrosis, a strong predictor of liver-related death (Neuschwander-Tetri 2014).

The FXR-SHP cascade is postulated to mediate the links between lipid and glucose metabolism (Zhang 2008, Cariou 2006, Rizzo 2006, Ma 2006, Shulman 2005).

OCA induces lipid uptake by mouse adipocyte cell line (3T3-L1) and primary human adipocytes, which correlate with reduced hepatic and circulating lipid levels, together with increased insulin sensitivity (Rizzo 2009, Rizzo 2006). Moreover, OCA significantly enhances adiponectin and leptin secretion by mouse and human adipocytes, which can enhance insulin sensitivity in peripheral tissues. Pancreatic beta cells express FXR messenger ribonucleic acid (mRNA) and protein, and OCA significantly enhances insulin secretion by mouse  $\beta$ -TC6 cells and human pancreatic islets (Rizzo 2009).

Collectively, these results indicate that OCA improves glycemia by increasing peripheral glucose uptake, enhancing glucose-stimulated insulin secretion, and inhibiting hepatic lipid synthesis and content while inducing lipid uptake by adipocytes (Adorini 2012, Mudaliar 2013).

# 5.4. Nonclinical Experience with Obeticholic Acid

Nonclinical studies have shown several potentially beneficial properties of FXR agonism in NASH, including

Effects of OCA on glycemic, metabolic, and cardiovascular properties

- FXR plays a role in bile acid homeostasis, metabolism, and clearance (Zhang 2008, Ma 2006, Cariou 2006).
- FXR controls glucose metabolism through regulation of gluconeogenesis and glycogenolysis in the liver, as well as regulation of peripheral insulin sensitivity in striated muscle and adipose tissue (Mudaliar 2013, Zhang 2006).
- In nonclinical models, FXR agonism is associated with beneficial effects on body weight and composition (Xu 2009, Fu 2004).
- The absence of endogenous intact FXR signaling results in dyslipidemia and a hepatic phenotype similar to NASH patients (Zhang 2008). Conversely, FXR agonists lower plasma TGs by repressing hepatic sterol regulatory element binding protein 1-c (Watanabe 2004) and increased hepatic fatty acid oxidation (Savkur 2005).
- In addition, OCA and other FXR agonists are anti-atherogenic and cardioprotective in animal models (Hartman 2009, Miyazaki-Anzai 2010).

## Anti-inflammatory and anti-fibrotic effects of OCA

• OCA exerts direct effects on serum-starved LX2 cells (an immortalized hepatic stellate cell line) to reduce the expression of key fibrotic genes (collagen I, alpha smooth muscle actin, transforming growth factor β-1 and matrix metalloproteinases; (Albanis 2005).

- In primary and cultured hepatocytes treated with pro-inflammatory mediators, OCA exerted direct effects to inhibit pro-inflammatory gene expression (eg, tumor necrosis factor-α [TNF-α], cyclooxygenase-2 [COX-2], and inducible nitric oxide synthase [iNOS]; (Wang 2008, Li 2007).
- FXR activation (with WAY-362450) reduced inflammatory cell infiltration and hepatic fibrosis in a mouse model of NASH (Zhang 2009).
- OCA improved portal hypertension in cirrhosis models (Mookerjee 2014).
- OCA inhibited gastrointestinal inflammation and preserves intestinal barrier function in models of inflammatory bowel diseases (Gadaleta 2011).

## Effects of OCA on diabetic nephropathy

- OCA ameliorates TG accumulation by modulating fatty acid synthesis and oxidation in a murine model of diet-induced obesity (Wang 2009)
- In the same murine model of diet-induced obesity, OCA improves proteinuria, prevents podocyte loss, mesangial expansion, accumulation of extracellular matrix proteins, and increased expression of pro-fibrotic growth factors and fibrosis markers, and reduces inflammation and oxidative stress (Wang 2009)
- In a murine model of diabetes, OCA improves renal injury by decreasing proteinuria, glomerulosclerosis, and tubulointerstitial fibrosis, and modulating renal lipid metabolism, macrophage infiltration, renal expression of SREBPs, pro-fibrotic growth factors, and oxidative stress enzymes (Wang 2010)

In summary, there is strong rationale to advance OCA for the treatment of NASH based on its FXR-mediated hepatoprotective properties and results indicating that OCA improves glycemia by increasing peripheral glucose uptake, enhances glucose-stimulated insulin secretion, and inhibits hepatic lipid synthesis and content while inducing lipid uptake by adipocytes.

# **5.5.** Clinical Experience with Obeticholic Acid

OCA is under investigation for the treatment of multiple chronic liver diseases, including the treatment of NASH, primary biliary cirrhosis (PBC, also known as primary biliary cholangitis [Beuers 2015a, Beuers 2015b, Beuers 2015c]), primary sclerosing cholangitis (PSC), and biliary atresia. The clinical development program for OCA includes the following 3 studies conducted using subjects with NAFLD or NASH:

• Study 747-203: A proof-of-concept, Phase 2 study in subjects with type 2 diabetes and NAFLD to evaluate the effects of OCA on insulin sensitivity (Mudaliar 2013)

• <u>FXR Ligand OCA in NASH Treatment (FLINT)</u>: A Phase 2 study conducted by the National Institute of Diabetes and Digestive and Kidney Diseases and the NASH CRN to evaluate the efficacy and safety of OCA in the treatment of NASH (Neuschwander-Tetri 2014)

• Study D8602001: A Phase 2 study conducted by Intercept's Asian development partner (Sumitomo Dainippon Pharma Co., Ltd) to evaluate the efficacy and safety of 3 doses of OCA versus placebo in NASH

Study 747-203 showed improved insulin sensitivity in subjects with type 2 diabetes and NAFLD, demonstrating the clinical relevance of the FXR agonist pathway and supporting the potential of OCA to treat NAFLD and/or NASH. With the exception of weight loss, OCA 25 mg appeared to be at least as effective as OCA 50 mg for the majority of endpoints evaluated.

The FLINT study demonstrated that OCA was superior to placebo in improving not only the key histologic features important in the underlying pathophysiology of the disease (inflammation, ballooning, steatosis), but notably that OCA was superior to placebo in improving fibrosis, a strong predictor of liver-related death. OCA treatment was also associated with improvement in markers of hepatocellular injury and some cardiometabolic features including weight and systolic blood pressure. Salutary effects on weight and blood pressure are important considerations since patients with NASH present with higher cardiovascular risk given the comorbidities of obesity and diabetes.

On average, LDL cholesterol demonstrated a significant increase in subjects treated with OCA compared to placebo; however, this increase was reversed and LDL cholesterol returned to below baseline levels in subjects who initiated statin therapy. The change in lipid profile, which was attenuated with continued treatment and reversed post-treatment, needs to be further investigated mechanistically and with respect to clinical management with standard of care statin therapy. With the exception of pruritus, which occurred more frequently in the OCA-treated subjects (23% OCA versus 6% placebo) and led to 1 discontinuation, the general adverse event (AE) profile was similar across both groups. There were 2 deaths in the FLINT study, both in OCA treatment groups (one from sepsis and congestive heart failure, and the other from cardiac ischemia or infarction (Neuschwander-Tetri 2014). The event of cardiac ischemia or infarction was assessed by the Investigator as possibly related to OCA while the event of sepsis was assessed as unrelated to OCA by the Investigator (Data on File).

Study D8602001 demonstrated a dose-dependent increase in the percentage of OCA-treated subjects compared to placebo subjects who achieved the primary endpoint (p = 0.053, not significant). The 40 mg OCA dose group achieved statistical significance for the primary endpoint compared to placebo (p = 0.0496). Dose-dependent trends not reaching statistical significance were also observed for several other pre-specified histologic endpoints, including the proportion of subjects with steatosis and inflammation improvement, ballooning resolution, and NASH resolution. In the completer analysis, similar dose-dependent effects were observed, with 51% of patients in the 40 mg dose group compared to 22% in the placebo group meeting the primary endpoint (p = 0.0061). With the exception of dose-dependent pruritus, OCA appeared to be generally safe and well tolerated. The number of pruritus-associated discontinuations were 0, 0, 2, and 5 subjects in the placebo, 10 mg, 20 mg, and 40 mg OCA groups, respectively. Changes in lipid parameters were directionally similar to those observed in the FLINT study.

No other meaningful differences in the rate of AEs between the OCA and placebo groups were noted.

Overall, the safety and efficacy profiles of OCA support a favorable benefit-risk ratio and demonstrate that OCA is a potentially important therapeutic option for patients with NASH, PBC, and other liver and gastrointestinal conditions. Pruritus is the most common dose-related AE associated with OCA treatment, especially in subjects with cholestasis. Other potential risks include liver toxicity and lipid profile abnormalities.

# 5.6. Rationale for Study Design, Doses of Investigational Product and Use of Atorvastatin

## 5.6.1. Rational for Study Design

As described in Section 5.1, the incidence of NASH is increasing and is likely to be the leading cause of liver transplant by 2020, highlighting the need for development of effective therapies that may improve steatohepatitis and resulting fibrosis, potentially delaying liver transplant or death. Given the atherosclerotic risk associated with elevations in LDL cholesterol, which are common in NASH, and also an observed effect of treatment with OCA, it is important to characterize the changes observed in circulating cholesterol associated with OCA treatment and the potential for management of those changes.

FXR has been shown to play an important role in lipid homeostasis and atherosclerosis with the potential to modulate circulating levels of both LDL and HDL cholesterol, which are components of cardiovascular prognosis in rodents (Gautier 2013, Zhang 2010, Nissen 2007). Similarly, the FLINT study demonstrated OCA-related changes in LDL and HDL cholesterol (Neuschwander-Tetri 2014). While the observed changes in LDL cholesterol in both rodents and humans run counter to changes that have been typically associated with improved cardiovascular health, animal data have consistently shown FXR agonism to be associated with reductions in atherosclerotic plaque formation. Rodent studies have shown that this anti-atherogenic effect with FXR agonism is possibly due to an increase in the hepatic clearance of excess cholesterol (Mencarelli 2009, Hartman 2009, Zhang 2010). It should be noted that the relevance of these findings to humans needs further evaluation due to differences in human and rodent lipid physiology.

In addition to cholesterol concentration, lipoprotein particle concentration and sizes have emerged as important factors in the evaluation of cardiovascular risk (Jeyarajah 2006). A recent Veterans Affairs study assessing LDL and HDL cholesterol concentrations, as well as particle size and numbers, in subjects treated with gemfibrozil demonstrated that these factors were stronger predictors of cardiovascular risk or benefit, respectively, than cholesterol concentrations (Otvos 2006). Consistently, examination of LDL and HDL cholesterol concentrations and particle concentration from the Framingham Offspring cohort (n = 3066), showed that LDL particle concentration was more predictive of cardiovascular risk (Cromwell 2007).

Given the complex role of FXR in lipid homeostasis, the observations of OCA on HDL and LDL concentrations in NAFLD and NASH, and the importance of evaluating the underlying function and composition of apolipoproteins, it is essential to evaluate the effect of OCA on these lipid-driven mechanisms of cardiovascular risk/benefit when considering OCA as a potential treatment for NASH. As such, this study, 747-209, will evaluate the effect of OCA on lipid

metabolism and the subsequent management of lipid changes with atorvastatin therapy. Evaluated parameters will include changes in cholesterol concentrations, lipoprotein particle size and number, apolipoprotein concentrations and the effects on reverse cholesterol transport in subjects with NASH.

# **5.6.2.** Rationale for Placebo Control Group

The use of a randomized placebo control will provide the best scientific evidence of safety and efficacy of OCA in NASH subjects. As there is no approved or proven pharmacologic therapy for NASH, the use of a placebo arm for comparative analysis is desired for robust analysis of efficacy and safety data. As the intent of the present study is to assess the effects of multiple doses of OCA and the subsequent addition of atorvastatin on cholesterol metabolism as well as the safety and tolerability of OCA in subjects with NASH, it is important to include a placebo control group to understand the relationship to OCA of any changes observed. In addition, the combination of OCA and atorvastatin (or any other statin) has not been previously evaluated in clinical studies; thus, the placebo control group, which will be treated with atorvastatin, will provide comparative information regarding the safety and tolerability of the OCA and atorvastatin combination compared to atorvastatin alone.

#### **5.6.3.** Rationale for OCA Doses

The selection of OCA doses for the present study (5 mg, 10 mg, and 25 mg) was guided by the available safety and tolerability data from randomized, double-blind, placebo-controlled Phase 2 and Phase 3 studies in subjects with NAFLD, NASH, and PBC as described in Section 5.5 above.

In Study 747-203, subjects with type 2 diabetes and NAFLD were treated with placebo, OCA 25 mg, or OCA 50 mg for 6 weeks. Although both doses were similarly efficacious, there were clinically significant increases in the LDLc levels in both OCA dose groups, with a significant reduction in HDL observed in the OCA 50 mg treatment group. Similarly, OCA was efficacious and well-tolerated in the subsequent, Phase 2, randomized, double-blind FLINT study, which evaluated OCA 25 mg and placebo in subjects with NASH over a period of 72 weeks. In this study, small but statistically significant changes in the levels of total cholesterol and LDLc levels (increase from Baseline), and HDL levels (decrease from Baseline) were observed with OCA treatment. Due to the similarity in efficacy and the observed lipoprotein changes in the two Phase 2 studies in subjects with NASH, OCA 25 mg will be the maximum dose in this study.

There was an increased incidence of mostly mild or moderate pruritus in OCA-treated subjects compared to placebo-treated subjects in the FLINT study. Pruritus was also the most common AE associated with OCA in PBC studies, and has been shown to be dose-related, warranting evaluation of lower doses as a potential strategy to improve tolerability. Phase 2 and Phase 3 studies evaluating OCA for the treatment of PBC have shown that the incidence and severity of pruritus with OCA treatment can be mitigated with lower OCA doses of 5 mg to 10 mg. Therefore, based on the therapeutic effect of 10 mg in PBC and to evaluate potential attenuation of the effect of OCA on pruritus and serum lipid levels, both 5 mg and 10 mg daily will be evaluated in the proposed NASH study in addition to the 25-mg dose.

#### **5.6.4.** Rationale for the Use of Atorvastatin

Subsequent to diet and lifestyle modification, statin therapy is recommended for the management of cholesterol to reduce cardiovascular risk globally (Perk 2012, NICE 2014, Stone 2014). Atorvastatin is one of the most commonly used statins worldwide (Jackevicius 2012). Historically, statin therapy has been contraindicated in subjects with elevations in liver aminotransferases. However, several studies have evaluated statin use in chronic liver diseases where cardiovascular risk is a significant concern and the consensus findings have not shown an increased risk of hepatotoxicity in subjects with elevated liver aminotransferases. Calderon et al reported that statin treatment is safe and can improve both liver aminotransferase levels and reduce cardiovascular morbidity (Calderon 2010, Tikkanen 2013, Athyros 2010).

The increase in LDL cholesterol levels in the OCA-treated NASH population observed in clinical studies may predispose these subjects to increased cardiovascular risk. Atorvastatin is one of the most widely prescribed statins for dyslipidemia in North America (Jackevicius 2012, Jackevicius 2013). The atorvastatin prescribing information suggests a starting dose of 10 mg, with dose adjustments every 2 to 4 weeks. In line with this recommendation, all subjects will be started at an atorvastatin dose of 10 mg at Week 4, titrating to 20 mg atorvastatin at Week 8 (if 10 mg daily is tolerated), and allowing for further dose adjustments at Week 12 based on clinical need and Investigator discretion.

In addition to mitigating the potential risk of statin use in this population by initiating treatment at the lowest indicated dose (10 mg once daily), subjects with excessive (>300 U/L) elevations in alanine aminotransferase (ALT), pre-existing cardiovascular disease, and those with elevated cardiovascular risk (eg, unstable hypertension) will be excluded. Finally, liver function, cholesterol levels, and vital signs will be monitored at all visits in this study, and investigational product will be withdrawn or its dosing interrupted in subjects who develop elevated levels of liver enzymes per protocol discontinuation criteria (see Section 8.4.1).

#### **5.6.4.1.** Rationale for Statin Withdrawal

The intent of this study is to assess the increase in LDL cholesterol with OCA and then to determine the extent to which this can be mitigated with appropriate use of statin therapy. Therefore, participating subjects need to either be statin-free or have washed off of their current statin therapy. Given the clear role of statins in reducing cardiovascular risk, it is imperative to minimize the potential risk associated with withdrawing statin therapy. These steps include minimizing the duration of statin withdrawal and exclusion of subjects for whom removal of statin therapy is of significant concern.

## Duration of statin withdrawal

A statin withdrawal period of 5 weeks was selected and is similar to other recent studies in statin-using patients where a 4-week washout period was employed (Teramoto 2012, Teramoto 2014). The extra week in the present study allows for the assessment of LDL levels after 4 weeks of washout, and based on prior studies, assumes levels of LDL to be stable after 4 weeks, and enables the stratification of subjects at randomization on Day 1 by this value.

Following randomization, subjects will be treated with OCA or placebo for 4 weeks prior to the introduction of atorvastatin. Based on data in healthy subjects, PBC, and NAFLD, 4 weeks is

sufficient to observe peak changes in LDL and HDL cholesterol due to OCA alone in most subjects.

Overall, statin therapy will be withheld from subjects for a maximum of 9 weeks: 5 weeks prior to randomization on Day 1 and 4 weeks following randomization. This duration of statin withdrawal is less than the combined withdrawal period used in the Teramoto et al study, which included a group of subjects who had statin therapy withheld for a total of 16 weeks (4 week washout period followed by 12 weeks of placebo treatment) (Teramoto 2014). There was no appreciable difference in the safety profile of these patients compared to those who had statin therapy reintroduced after the washout period. Further support for the minimal impact of short-term discontinuation of statins is seen in follow-up analyses of the Treating to New Target study which showed that even in patients with stable coronary artery disease, that a 6-week interruption of statin therapy did not acutely impact cardiac events (McGowan 2004).

### Exclusion of subjects at elevated risk

Subjects where the removal of a statin would be considered to be clinically concerning are excluded from participation in this study. At risk subjects include subjects with existing cardiovascular disease (including but not limited to stable or unstable angina, previous myocardial infarction or stroke or a previous peripheral or coronary revascularization procedure), significant dyslipidemia (as defined by LDLc  $\geq$ 190 mg/dL) despite the use of statin therapy, unstable hypertension, and familial hypercholesterolemia.

Safety monitoring during the off-statin period

All subjects will have frequent safety assessments prior to and following the reintroduction of statin therapy. Following Screening Visit 1, subjects will have 4 visits to the study site over the 9-week period prior to initiation of atorvastatin: Screening Visit 2/Week -1, Randomization/Day 1, Week 2 and Week 4. During these visits AEs, vital signs, and safety labs will be assessed and monitored by the site staff.

#### **5.6.5.** Rationale for Duration of Treatment

In the clinical studies where healthy subjects and subjects with PBC were treated with OCA, changes in cholesterol were evident by 2 weeks of treatment. Accordingly, the effect of OCA on lipoprotein metabolism, prior to the introduction of atorvastatin, will be assessed at 2 and 4 weeks of treatment to evaluate the change in these parameters and the effect of sustained treatment with OCA; all subjects will then initiate atorvastatin therapy, in addition to their blinded treatment, and the effect on lipoprotein metabolism will be evaluated over an additional 12 weeks. The total duration of the double-blind phase of the study is 16 weeks, which is sufficient to evaluate the effect of atorvastatin on the OCA treatment-induced alterations in the lipoprotein profile of statin-naïve and statin-washed out NASH subjects.

Following the double-blind phase, subjects may volunteer to continue in a 2-year open-label long-term safety extension (LTSE) during which all subjects will receive OCA. During the LTSE, LDL cholesterol will be managed as clinically indicated. The LTSE will evaluate the long-term safety of OCA and atorvastatin treatment and the effect of OCA and atorvastatin on histological markers of NASH.

# 5.6.6. Rationale for Timing of Unblinding Process and Implications in LTSE

As Study 747-209 is a randomized, double-blind study, the double-blind data will not be unblinded until all double-blind data are final and the database is locked. Accordingly, all subjects continuing in the LTSE, Investigators, and the Sponsor will remain blinded to subjects' double-blind treatment regimen. Subjects who were receiving placebo or 5 mg OCA in the double-blind phase will be randomized to receive either OCA 10 mg or OCA 25 mg in the LTSE. Subjects who were receiving OCA 10 mg or OCA 25 mg in the double-blind phase will continue on the same dose throughout the LTSE. Using this approach, blinding of the trial will be maintained.

# 5.7. Summary of Known Potential Risks with Investigational Product

The primary AE shown to be related to OCA is pruritus. Pruritus has also been observed in clinical studies with OCA in other indications, as well as in healthy subjects, with the highest frequency observed in subjects with PBC.

An increase in liver enzymes and hepatic AEs, including jaundice, were observed in subjects with liver disease at OCA doses between 10 mg and 50 mg. Elevated liver enzymes were observed in healthy subjects who were treated at doses  $\geq$ 100 mg in Phase 1, multiple-dose studies; however, these elevations were only considered to be of clinical concern at the maximum dose of 250 mg daily.

Changes in lipid profiles have also been observed with OCA dosing, including a decrease in HDL cholesterol and an increase in LDL cholesterol. The clinical significance of these lipid findings remains unclear and is being studied further. HDL levels have generally remained within normal limits in subjects treated with OCA. While LDLc levels increased with OCA treatment, the changes were modest, and trended toward baseline values with continued treatment through to 72 weeks.

Refer to the Investigator's Brochure (IB) for additional information regarding the known potential risks with the investigational product.

# 5.8. Summary of Known Potential Risks with Atorvastatin

Muscle complaints are the most frequent adverse reports among patients treated with statins with the most severe side effects including myopathy and rhabdomyolysis. The Statin Muscle Safety Task Force (Rosenson 2014) has provided a classification of the spectrum of statin-associated muscle AEs that may be seen in clinical practice and can be used in characterizing reports of muscle-related events.

- a. Myalgia unexplained muscle discomfort often described as "flu-like" symptoms
  - Muscle aches
  - Muscle soreness
  - Muscle stiffness
  - Muscle tenderness
  - Muscle cramps with or shortly after exercise (not nocturnal cramping)
b. Myopathy – muscle weakness (not attributed to pain and not necessarily associated with elevated CPK)

- c. Myositis muscle inflammation
- d. Myonecrosis muscle enzyme elevations or hyperCPKemia
  - Mild >3x baseline or ULN
  - Moderate >10x baseline or ULN
  - Severe >50x baseline or ULN
- e. Clinical Rhabdomyolysis Myonecrosis with myoglobinuria or acute renal failure (increase in serum creatinine ≥0.5 mg/dL

There is no evidence that these muscle-related AEs are a continuum beginning with myalgia and progressing to more severe manifestations of myopathy; rather events occur independent of each other. Myalgia events, with frequencies ranging from 1% to 5% in clinical trials to 11% to 29% in observational cohorts, typically occur within 1 month of statin initiation and resolve within 2 weeks of statin cessation (Rosenson 2014). Retrospective analyses have suggested that patients who discontinue statins due to intolerance are able to tolerate statins long-term following re-challenge (Zhang 2013, Mampuya 2013).

Historically, statins have been associated with biochemical abnormalities of liver function, but available data suggest that increases in liver transaminases associated with statins are asymptomatic and generally reversible (Desai 2014). In the absence of liver disease, US guidelines (Stone 2013) recommend that baseline transaminase levels should be checked before initiating statin therapy and subsequent testing should only be done in the presence of symptoms suggestive of hepatic disease. As this study is being conducted in subjects with confirmed NASH, liver enzymes will be frequently monitored and Section 8.4.1.3, Section 8.4.2.2, and Appendix B provide detailed guidance for handling elevated liver biochemistry values.

Statins modestly increase the risk of type 2 diabetes mellitus in individuals with risk factors for diabetes. Individuals receiving statin therapy should be evaluated for new-onset diabetes according to the current diabetes screening guidelines (American Diabetes Association 2013).

Confusion and memory loss have been reported with statins, but medical evidence supporting a causal effect is weak or nonexistent (Simic 2015). However, any reports of cognitive events should be appropriately evaluated, particularly in individuals whose symptoms persist despite statin discontinuation.

In this study, any AEs (including signs and symptoms described above) regardless of relationship to investigational product or study medication, must be documented appropriately (see Section 12).

If treatment with statins is initiated, women of childbearing potential must be informed that statin use is contraindicated during pregnancy. Methods of contraception should be reviewed and modified, if necessary, to ensure highly effective methods with failure rates <1% per year, such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or history of vasectomy of partner are used.

## 6. STUDY OBJECTIVES AND PURPOSE

# 6.1. Primary Objective

The primary objective of the study is:

• To evaluate the effect of OCA on LDL metabolism in subjects with biopsy-confirmed NASH and to assess the ability of atorvastatin to modulate this effect

# **6.2.** Secondary Objectives

The secondary objectives of the study are:

- To evaluate the safety and tolerability of OCA alone and in combination with atorvastatin therapy in subjects with biopsy-confirmed NASH
- To evaluate the effect of OCA with and without atorvastatin therapy, on
  - HDL, VLDL, TGs, total cholesterol, and apolipoprotein concentrations
  - Components of the reverse cholesterol transport pathway

# **6.3.** Exploratory Objectives

The exploratory objectives of the study are:

- To evaluate the effect of OCA on
  - Liver biochemistry, inflammation, and apoptosis
  - Markers of glucose metabolism including C-peptide, insulin, fasting plasma glucose, hemoglobin-specific A1c fraction (HbA1c), homeostatic model assessment-beta-cell function (HOMA-β), and homeostatic model assessment – insulin resistance (HOMA-IR)
  - Anthropometric measures including height (measured at Screening Visit 1 only), weight, and waist and hip circumference measurements; and body mass index (BMI), and waist-to-hip ratio calculations
  - Cardiovascular risk scores (eg, Framingham Risk Score [FRS] and Reynolds score)
  - To evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of OCA and its conjugates
  - To evaluate the bioanalytical concentrations of atorvastatin and its metabolites
  - To evaluate improvement in noninvasive-radiological assessment of fibrosis via transient elastography (TE; at sites where available)

## 7. INVESTIGATIONAL PLAN

# 7.1. Overall Study Design

This Phase 2, double-blind, randomized, placebo-controlled, multicenter study, with an open-label LTSE, will evaluate the effect of OCA, and the subsequent addition of statin therapy, on lipoprotein metabolism in subjects with NASH with fibrosis stage 1 to 4, but no evidence of hepatic decompensation. Approximately 80 subjects with histological evidence of definite or probable NASH, who meet all inclusion and none of the exclusion criteria will be enrolled in the study. The histological evidence of definite or probable NASH will be based on the central read of a liver biopsy obtained no more than 1 year prior to randomization and a nonalcoholic fatty liver disease activity score (NAS) of 4 or greater. Subjects not using statin therapy (ie, statin-free) and statin-treated subjects may be enrolled. Statin-treated subjects will be required to stop statin treatment (after signing informed consent) for up to 5 weeks, including a 4-week statin washout period, prior to Randomization/Day 1.

## **Screening Period:**

Subjects will have a screening period of up to 5 weeks prior to Randomization/Day 1.

Subjects using statins within 30 days of the initial Screening Visit (Screening Visit 1) are required to stop statin therapy immediately following this initial visit and must undergo a 4-week statin washout period prior to Screening Visit 2. At Screening Visit 2 these subjects will have a pre-randomization visit for assessment of their fasting LDL cholesterol levels. Subjects with fasting LDL cholesterol values >200 mg/dL at Screening Visit 2 will be excluded from the study and their dyslipidemia should be managed according to standard of care.

Subjects who are not using statin therapy at Screening Visit 1 are required to provide a fasting blood sample at Screening Visit 2, which can occur at any time prior to randomization but after signing of the ICF. Statin free subjects with fasting LDL cholesterol values >200 mg/dL at either Screening Visit will be excluded from the study and should be managed according to standard of care.

#### **Double-Blind Phase:**

At the Randomization (Day 1) Visit, subjects will be randomized in a 1:1:1:1 ratio to receive OCA 5 mg, OCA 10 mg, OCA 25 mg, or placebo, orally, once daily, for 16 weeks. Randomization will be stratified by the pre-randomization fasted serum LDL cholesterol concentration (≤125 mg/dL or >125 mg/dL) and baseline fibrosis stage (stage 1, 2 or stage 3, 4).

At the Week 4 Visit, all subjects will initiate treatment with atorvastatin at a dose of 10 mg once daily. At the Week 8 Visit, atorvastatin will be increased to 20 mg once daily (if 10 mg daily is tolerated), and continued for an additional 4 weeks. After 4 weeks of treatment at 20 mg, the atorvastatin dose may be titrated (up or down) as clinically indicated. The final visit during the double-blind phase will occur at Week 16, after which subjects may continue into the open-label LTSE.

Subjects who discontinue investigational product or atorvastatin during the double-blind phase are still expected to attend scheduled study visits and are to be followed through the Week 16 Visit.

Subjects who discontinue atorvastatin during the double-blind phase are eligible to continue OCA during the double-blind phase and enroll into the LTSE at the discretion of the Investigator, provided they continue to meet the LDLc cutoff of exclusion criteria #4 (ie, LDLc <200 mg/dL).

#### LTSE Phase:

During the LTSE phase, all subjects will be treated with open-label OCA 10 mg or OCA 25 mg. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will be randomized in a 1:1 ratio to receive OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg or OCA 25 mg during the double-blind phase will continue on the same dose throughout the LTSE. In the event of OCA-related tolerability concerns, the Investigator may refer to the IB for possible treatment options. Subjects may continue, discontinue, or modify the atorvastatin therapy as clinically indicated.

## 7.1.1. Study Design

Figure 1: Study Design Schematic



LTSE: long-term safety extension; Wk = week Note: Statin therapy refers to atorvastatin.

 $\Delta$  = Telephone Safety Contact at Week 6, Week 10, and Week 14

# 7.1.2. Schedule of Study Procedures

Table 1: Schedule of Study Procedures: Double-Blind Period

| Study Visits | Screening<br>Visit 1 <sup>a</sup> | Screening<br>Visit 2 <sup>b</sup> | Randomi-<br>zation/ Day 1 | Wk 2 | Wk 4 | Wk 6<br>(Contact) | Wk8 | Wk 10<br>(Contact) | Wk 12 | Wk 14<br>(Contact) | Wk 16/<br>LTSE Day 1 | ET/<br>EOS <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | -5 to -1 | -1 to 1 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | |
| Visit Window (Days) | -35 to -7 | -7 to -1 | | ±4 | ±4 | ±4 | ±4 | ±4 | ±4 | ±4 | ±4 | ±7° |
| STUDY PROCEDURES | STUDY PROCEDURES | | | | | | | | | | | |
| Fast ≥8 h Prior to Visit | | X | X | X | X | | X | | X | | X | X |
| Informed Consent | X | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | X | X | | | | | | | | | |
| Physical Exam | X | | | | | | | | | | X | X |
| Vital Signs <sup>d</sup> | X | | X | X | X | | X | | X | | X | X |
| Anthropometric Measures <sup>e</sup> | X | | X | X | X | | X | | X | | X | X |
| 12- Lead<br>Electrocardiogram | X | | X | | | | | | | | X | X |
| AUDIT Alcohol Intake<br>Questionnaire | X | | X | | | | | | | | X | X |
| Liver Biopsy <sup>f</sup> | X | | | | | | | | | | | |
| Transient Elastography <sup>g</sup> | X | X | X | | | | | | | | X | X |
| AEs <sup>h</sup> | X <sup>h</sup> | X <sup>h</sup> | X | X | X | X | X | X | X | X | X | X |
| Prior and Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization/Treatment<br>Assigned <sup>i</sup> | | | Xi | | | | | | | | Xi | |
| Dispense/Administer<br>Investigational Product <sup>k</sup> | | | X | X | X | | X | | X | | X <sup>j</sup> | |
| Dispense/Administer<br>Open-Label Atorvastatin <sup>k</sup> | | | | | X | | X | | X | | X <sup>j</sup> | |

**Table 1: Schedule of Study Procedures: Double-Blind Period (Continued)** 

| Study Visits | Screening<br>Visit 1 <sup>a</sup> | Screening<br>Visit 2/<br>Wk -1 <sup>b</sup> | Randomi-<br>zation/<br>Day 1 | Wk 2 | Wk 4 | Wk 6<br>(Contact) | Wk8 | Wk 10<br>(Contact) | Wk<br>12 | Wk 14<br>(Contact) | Wk 16/<br>LTSE<br>Day 1 | ET/<br>EOS <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Collect Bottles/Investigational Product Accountability/Compliance | | | | X | X | X | X | X | X | X | X | X |
| Collect Bottles/Atorvastatin<br>Accountability/Compliance | | | | | | | X | X | X | X | X | X |
| CLINICAL LABORATOR | Y EVALUAT | TIONSk | | | | | | | | | | |
| Hepatitis B Virus and<br>Hepatitis C Virus Tests | X | | | | | | | | | | | |
| Serum Chemistry <sup>l, m</sup><br>/Hematology/ Coagulation<br>Parameters | X | X | X | X | X | | X | | X | | X | X |
| Lipoprotein Analyses <sup>n</sup> | | | X | X | X | | X | | X | | X | X |
| Reverse Cholesterol<br>Transport Analytes <sup>o</sup> | | | X | X | X | | X | | X | | X | X |
| PD Assessments | | | X | | X | | X | | X | | X | X |
| Markers of Inflammation,<br>Fibrosis, and Apoptosis | | | X | | X | | X | | X | | X | X |
| Vitamin D | | | X | | X | | X | | X | | X | X |
| Markers of Glucose<br>Metabolism Including<br>C-peptide, Insulin, Fasting<br>Plasma Glucose, and<br>HbA1c <sup>p</sup> | | | X | | X | | X | | X | | X | X |
| Thyroid Function Tests:<br>T3, T4, and TSH | | | X | | | | | | | | X | X |
| Urinalysis | X | | X | | | | | | | | X | X |
| Pregnancy Test <sup>q</sup> | Xq | | X | X | X | | X | | X | | X | X |
| Blood Sample for Future<br>Exploratory Analysis <sup>r</sup> | | | X | | | | X | | | | X | X |
| PK Assessments <sup>s</sup> | | | Xs | | | | | | | | Xs | |

AE = adverse event; AUDIT = Alcohol Use Disorders Identification Test;  $\beta$ -hCG = beta human chorionic gonadotropin; BMI = body mass index; CPK = creatine phosphokinase; EOS = End of Study; ET = Early Termination; HbA1c = hemoglobin-specific A1c fraction; hs-CRP = high-sensitivity C-reactive protein; PD = pharmacodynamics; PK = pharmacokinetics; T3 = triiodothyronine; T4 = thyroxine; TSH = thyroid-stimulating hormone; Wk = Week Note: No study-related procedures, including Screening procedures, will be performed prior to obtaining informed consent from the subject. Historical procedures (eg, liver biopsy samples collected, FibroScan) completed as part of standard of care, may be used for screening analysis if collected within the allowed windows specified in the protocol.

- <sup>a</sup> Subjects using statins within 30 days of Screening are required to stop administering statin therapy after Screening Visit 1, and must complete a 4-week statin washout prior to performing assessments at Screening Visit 2.
- b Screening Visit 2 is required for all subjects. All subjects must have been fasting for at least 8 hours prior to the visit. The Randomization/Day 1 Visit may occur as soon as screening labs are available and eligibility is confirmed for all subjects. For subjects undergoing a 4-week washout period, Screening Visit 2 may occur on day 28 (±1) day of the washout period. For subjects not taking statins at Screening Visit 1, Screening Visit 2 can occur at any time within 28 days after Screening Visit 1. All Screening assessments must be completed ≤35 days prior to the Randomization/Day 1 Visit.
- <sup>c</sup> The ET Visit will occur as soon as possible upon study discontinuation and as near as possible to last dose taken. The EOS Visit will occur ±1 week (7 days) relative to the EOS date announced by the Sponsor.
- <sup>d</sup> Sitting heart rate, blood pressure, body temperature, and respiratory rate.
- e Weight, waist and hip circumference (and height at Screening Visit 1). BMI and waist-to-hip ratio will be calculated via electronic data capture (EDC).
- f Liver biopsy will be performed to histologically confirm NASH only if slides from historic biopsy (within 1 year of Day 1) are not available. A central reader designated by the Sponsor will perform all biopsy scoring; the results of which must be available prior to randomization on Day 1.
- Transient elastography (TE) will be conducted at selected trial sites where the FibroScan® TE device is available. TE is scheduled for Screening Visit 1; however, it may be performed any time after Screening Visit 1 and prior to randomization. In addition, if TE has been done within 3 months of Day 1 and a report/adequate data are available, a pretreatment TE at Day 1 is not required.
- <sup>h</sup> AEs occurring after the signing of the informed consent form (ICF) must be entered on the AE eCRF.
- <sup>1</sup> Only those subjects who were statin naive at Screening or who have successfully completed the washout period and meet all other inclusion criteria, and none of the exclusion criteria, may be randomized. Subjects randomized to placebo or OCA 5 mg during the double-blind period will be randomized to OCA 10 or 25 mg during the LTSE.
- <sup>j</sup> Only applies to subjects continuing in LTSE.
- <sup>k</sup> Blood samples for all analyses will be collected predose (before administering investigational product or atorvastatin) on indicated visit days.
- <sup>1</sup> CPK will be assessed in all subjects at Screening Visit 2 and as clinically indicated, including anytime myopathy is suspected.
- <sup>m</sup> Serum chemistry will include a basic lipid panel and also liver biochemistry panel (see Table 10).
- <sup>n</sup> Serum and plasma samples will be collected for lipoprotein analysis, which will include cholesterol concentration in LDL, HDL, and VLDL, their particle concentration and sizes; concentrations of apolipoprotein (Apo)A1, ApoB, ApoE, ApoCII, ApoCIII and Lp(a); and proprotein convertase subtilisin/kexin type 9 (PCSK9).
- ° Reverse cholesterol transport analysis will include following analytes: Pre-β1 HDL concentration, macrophage cholesterol efflux, lecithin cholesterol acyltransferase activity, and cholesterol ester transfer protein activity.
- <sup>p</sup> The homeostatic model assessment–beta-cell function (HOMA-β) and homeostatic model assessment insulin resistance (HOMA-IR) indexes will be calculated using fasting plasma glucose and serum insulin values.
- <sup>q</sup> Serum pregnancy test will be administered if urine-based β-hCG pregnancy test is positive. Screening pregnancy tests will be serum-based tests.
- <sup>r</sup> Includes markers of cardiovascular risk (adiponectin, plasminogen activator inhibitor-[(PAI-1], and B-type natriuretic peptide [BNP]).
- Shall selected investigational sites, subjects will have the option to provide blood samples for measurement of PK for OCA (Day 1 and Week 16), and for atorvastatin (Week 16). PK samples will be collected within 30 minutes prior to dosing and again at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until the 1 hour sample is collected.

Table 2: Schedule of Study Procedures: LTSE

| | | Annual Schedule (Year 1 through Study Termination) <sup>b</sup> | | | | |
|---|---|---|---|---|---|---|
| Study Visits | Month 1 <sup>a</sup> | Month 3,<br>Month 15 | Month 6,<br>Month 18 | Month 9,<br>Month 21 | Month 12 | EOS/ET <sup>e</sup> |
| Visit Windows (weeks) | ±1 | ±1 | ±1 | ±1 | ±1 | ±1/ N/A <sup>c</sup> |
| STUDY PROCEDURES | | | | | · | |
| Fast ≥8 h Prior to Visit | X | X | X | X | X | X |
| Physical Exam | | X | | | X | X |
| 12-Lead Electrocardiogram | | X | X | X | X | X |
| Vital Signs <sup>d</sup> | X | X | X | X | X | X |
| Anthropometric Measures <sup>e</sup> | | X | X | X | X | X |
| AUDIT Alcohol Intake Questionnaire | | | X | | X | X |
| AEs | X | X | X | X | X | X |
| Prior and Concomitant Medications | X | X | X | X | X | X |
| Transient Elastography <sup>f</sup> | | | | | X | X |
| Dispense/Administer Investigational Productg | | X | X | X | X | |
| Dispense/Administer Atorvastating,h,i | | X | X | X | X | |
| Collect Bottles/Investigational Product Accountability/Compliance | X | X | X | X | X | X |
| Collect Bottles/Atorvastatin Accountability/Compliance | X | X | X | X | X | X |
| LABORATORY EVALUATIONS <sup>g</sup> | | | | | | |
| Serum Chemistry <sup>j,k</sup> /Hematology/ Coagulation Parameters | X | X | X | X | X | X |
| Lipoprotein Analyses <sup>1</sup> | | X | X | X | X | X |
| Reverse Cholesterol Transport Analysis <sup>m</sup> | | | X | | X | X |
| PD Assessments | | X | X | X | X | X |
| Markers of Inflammation, Fibrosis, and Apoptosis | | X | X | X | X | X |
| Vitamin D | | X | X | X | X | X |
| Markers of Glucose Metabolism Including C-peptide,<br>Insulin, Fasting Plasma Glucose, HbA1c <sup>n</sup> | X | X | X | X | X | X |
| Thyroid Function Tests: T3, T4, and TSH | | | | | X | X |
| Urinalysis | | | | | X | X |
| Urine Based β-hCG Pregnancy Test <sup>o</sup> | X | X | X | X | X | X |
| Blood Sample for Future Exploratory Analysis <sup>p</sup> | | | | | X | X |

AE = adverse event; AUDIT = Alcohol Use Disorders Identification Test;  $\beta$ -hCG = beta human chorionic gonadotropin; BMI = body mass index; CPK = creatine phosphokinase; EOS = End of Study; ET = Early Termination; HbA1c = hemoglobin-specific A1c fraction; PD = pharmacodynamics; T3 = triiodothyronine; T4 = thyroxine; TSH = thyroid-stimulating hormone

- <sup>a</sup> The first visit after start of LTSE (Month 1 Visit) is relative to Week 16 Visit of the double-blind phase (LTSE Day 1 Visit).
- <sup>b</sup> After the Month 12 Visit, the procedures will be performed as listed for Month 3, Month 6, and Month 9 visits (at 15 months, 18 months, and 21 months, respectively, into the LTSE).
- <sup>c</sup> The ET Visit will occur as soon as possible upon study discontinuation and as near as possible to last dose taken. The EOS Visit will occur ±1 week (7 days) relative to the EOS date announced by the Sponsor.
- <sup>d</sup> Sitting heart rate, blood pressure, body temperature, and respiratory rate.
- <sup>e</sup> Weight, waist and hip circumference. BMI and waist-to-hip ratio will be calculated via electronic data capture (EDC).
- f Transient elastography (TE) will be conducted during the LTSE at selected trial sites where the FibroScan® TE device is available.
- <sup>g</sup> Blood samples for all analyses will be collected predose (before administering investigational product) on indicated visit days.
- <sup>h</sup> Atorvastatin may be continued or subjects may change or discontinue statins as clinically indicated.
- <sup>i</sup> **NOTE**: Any time atorvastatin is up-titrated or re-initiated, a telephone safety contact must be conducted to assess AEs, concomitant medications, and atorvastatin compliance.
- <sup>j</sup> CPK will be assessed in all subjects only as clinically indicated, including anytime myopathy is suspected, in subjects taking statins.
- <sup>k</sup> Serum chemistry will include a basic lipid panel and liver biochemistry panel (see Table 10).
- <sup>1</sup> Serum samples will be collected for lipoprotein analyses, which will include cholesterol concentration in LDL, HDL, and VLDL, their particle concentration and sizes; concentrations of apolipoprotein (Apo)A1, ApoB, ApoE, ApoCII, ApoCIII and Lp(a); and proprotein convertase subtilisin/kexin type 9 (PCSK9).
- m Reverse cholesterol transport analysis will include following analytes: Pre-β1 HDL concentration, macrophage cholesterol efflux, lecithin cholesterol acyltransferase activity, and cholesterol ester transfer protein activity.
- $^{n}$  The homeostatic model assessment-beta-cell function (HOMA- $\beta$ ) and homeostasis model assessment insulin resistance (HOMA-IR) indexes will be calculated using fasting plasma glucose and serum insulin values.
- $^{\circ}$  Serum pregnancy test will be administered if urine-based  $\beta$ -hCG pregnancy test is positive.
- <sup>p</sup> Blood sample for future exploratory analysis, including markers of cardiovascular risk (adiponectin, plasminogen activator inhibitor-[(PAI-1], and B-type natriuretic peptide [BNP]).

## 7.1.3. Study Duration

The overall study duration is up to 125 weeks including a Screening period of up to 5 weeks (depending on current statin use), a 16-week double-blind treatment phase, and a 2-year, open-label LTSE. The LTSE may be terminated earlier by the Sponsor if OCA becomes commercially available, or for other reasons as described in Section 8.4.3.

# 7.2. Number of Subjects

Approximately 80 subjects who meet the eligibility criteria, including biopsy-confirmed NASH and evidence of liver fibrosis, but no hepatic decompensation, will be included in this study. A maximum of 30% of subjects will have stage 4 fibrosis.

# 7.3. Treatment Assignment

Eligible subjects will be randomized into 4 groups in a 1:1:11 ratio to receive OCA 5 mg, OCA 10 mg, OCA 25 mg, or placebo during the double-blind phase of the study. Randomization will be stratified by LDL concentration (fasting serum LDL cholesterol at Screening Visit 2; ≤125 mg/dL or >125 mg/dL) and baseline fibrosis stage (stage 1, 2 or stage 3, 4). All subjects will also receive atorvastatin starting at Week 4 at 10 mg daily, escalating to 20 mg at Week 8 (if 10 mg daily is tolerated), with further dose adjustments to be performed as clinically indicated at Week 12, and throughout the LTSE phase. Subjects will receive open-label OCA 10 mg or OCA 25 mg during the LTSE depending on their double-blind randomized dose (see Section 7.1). The study design schematic is shown in Figure 1.

# 7.4. Dose Adjustment Criteria

# 7.4.1. Investigational Product Dose Adjustments

Dose adjustments of investigational product are not permitted during the double-blind phase. Please refer to Section 8.4.4 for instructions regarding subject withdrawal if investigational product is discontinued.

During the LTSE phase, all subjects will be treated with open-label OCA 10 mg or 25 mg. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will be re-randomized in a 1:1 ratio through IWRS to OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg will continue to receive OCA 10 mg throughout the LTSE. Subjects randomized to OCA 25 mg will continue to receive OCA 25 mg throughout the LTSE. Subjects may continue with atorvastatin therapy as clinically indicated.

## 7.4.2. Atorvastatin Dose Adjustments

For all subjects, atorvastatin therapy will be initiated at a dose of 10 mg at Week 4. At Week 8 the dose will be increased to 20 mg (if 10 mg daily is tolerated), and following the Week 12 Visit, the dose can be adjusted to manage cholesterol as clinically indicated (Section 9 and Appendix A). During the LTSE, subjects may continue with atorvastatin therapy as clinically indicated.

If at any time during the double-blind or LTSE phases, serum chemistry results indicate LDLc<40 mg/dL, the subject should be brought back to the site within 1 to 2 weeks after the first result is obtained for an unscheduled (repeat) laboratory assessment. If LDLc<40 mg/dL is obtained on 2 consecutive visits, the subject may discontinue or reduce the dose of atorvastatin.

Subjects may also interrupt or discontinue atorvastatin due to tolerability issues including muscle-related symptoms (Section 5.8) and abnormal liver biochemistry. Any muscle-related complaints should be assessed per the ACC/AHA Guidelines (Appendix A) and statin dose adjusted accordingly:

- To avoid unnecessary discontinuation of statins, obtain a history of prior or current muscle symptoms to establish a baseline prior to initiation of statin therapy.
- If mild to moderate muscle symptoms develop during statin therapy:
  - Discontinue the statin until symptoms can be evaluated.
  - Evaluate the patient for other conditions that might increase the risk for muscle symptoms.
  - If muscle symptoms resolve, and if no contraindication exists, re-challenge the subject with the same or a reduced dose of atorvastatin to establish a causal relationship between the muscle symptoms and statin therapy.
  - Once a low dose statin is tolerated, the dose may be gradually increased as tolerated and clinically indicated.
  - If after 2 months without statin treatment, muscle symptoms or elevated CPK levels do not completely resolve, consider other causes of muscle symptoms.
  - If persistent muscle symptoms are determined to arise from a condition unrelated to statin therapy, or if the predisposing condition has been treated, resume statin therapy at the original dose.
- If unexplained severe muscle symptoms or fatigue develop during statin therapy, discontinue the statin and address the possibility of rhabdomyolysis by evaluating CPK and serum creatinine, and performing urinalysis for myoglobinuria.

Elevations in liver biochemistry should be monitored per protocol subject withdrawal criteria (Section 8.4 and Appendix B).

Subjects who discontinue atorvastatin may continue on investigational product through the double-blind and LTSE phases, as deemed appropriate by the Investigator and Medical Monitor, and provided they continue to meet exclusion criteria #4 (LDLc <200 mg/dL).

#### 7.4.3. Safety Criteria for Adjustment or Stopping of Doses of Investigational Product

The Data Monitoring Committee (DMC) will review safety data from this study as well as other ongoing OCA studies on a periodic basis (Section 13.8). Adjustments to or discontinuation of treatment may be considered based on DMC evaluation of OCA safety and tolerability. The criteria for study termination are described in Section 7.5.

# 7.5. Criteria for Study Termination

The Sponsor reserves the right to terminate the study at any time. It is normal procedure to review the emerging clinical and safety data. As a result of such a review or a recommendation by the DMC, it may be necessary to stop the study before all subjects have completed the study. In addition, the Sponsor may terminate the study at an investigational site, at any time (eg, Good Clinical Practice [GCP] noncompliance, poorly performing sites, as determined by the number of subjects enrolled or the quality of the study data).

The Investigator and/or the Sponsor (or designee) must notify the Institutional Review Board/Independent Ethics Committee (IRB/IEC) of discontinuation of a site or the study and the reason(s) for doing so.

Investigators will be informed by the Sponsor as to when the final study visit is to be completed, and should then schedule all subjects for the End of Study (EOS) or Early Termination (ET) Visit.

#### 8. SELECTION AND WITHDRAWAL OF SUBJECTS

# 8.1. Subject Population

Approximately 80 subjects with biopsy-confirmed NASH without evidence of hepatic decompensation who meet eligibility criteria will be enrolled at approximately 30 investigational sites in the US. Prospective subjects will be identified primarily from the hospital and/or physician's database of patients with NASH, or may be referred from other physicians. Subjects may self-refer to an Investigator if they become aware of the study through local, national, or international NASH patient societies, forums, or networks. Subjects will be selected according to the inclusion and exclusion criteria below.

# 8.2. Subject Inclusion Criteria

Subjects must satisfy all of the following criteria to be eligible for enrollment:

- 1. Age  $\geq$ 18 years of age
- 2. Histologic evidence of NASH, as assessed by central reading of a liver biopsy obtained no more than 1 year prior to randomization, defined by the presence of all 3 key histological features of NASH with a score of at least 1 for each and a combined score of 4 or greater out of a possible 8 points according to NASH CRN criteria.
- 3. Histologic evidence of fibrosis stage 1 to stage 4 (as defined by NASH CRN scoring of fibrosis) without any evidence of hepatic decompensation.
- 4. If subject has type 2 diabetes, is on stable dose of anti-diabetic medication (except thiazolidinediones [TZDs]) for ≥3 months prior to Day 1.
- 5. Is either not taking or is on stable doses of TZDs and/or Vitamin E for ≥6 months prior to Day 1
- 6. Contraception: Female subjects of childbearing potential must use ≥1 effective method of contraception during the study and until 30 days following the last dose of

investigational product. Effective methods of contraception are considered to be those listed below.

- Barrier method, ie, condom (male or female) with spermicide or diaphragm with spermicide
- Intrauterine device
- Vasectomy (partner)
- Hormonal (eg, contraceptive pill, patch, intramuscular implant or injection)
- Abstinence (defined as refraining from heterosexual intercourse).
- 7. Must provide written informed consent and agree to comply with the study protocol, including adherence to protocol-described statin withdrawal and statin therapy.

# 8.3. Subject Exclusion Criteria

Subjects who satisfy any of the following exclusion criteria will be ineligible for enrollment:

- 1. Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to Screening Visit 1 (significant alcohol consumption is defined as more than 2 units/day in females and more than 4 units/day in males, on average).
- 2. Prior intolerance to treatment with atorvastatin or other 3-hydroxy-3-methyl-glutaryl (HMG) Coenzyme A reductase inhibitors (including but not limited to rhabdomyolysis).
- 3. LDLc ≥190 mg/dL and already on statin therapy at Screening Visit 1.
- 4. LDL cholesterol >200 mg/dL at any Screening Visit in subjects who are not on statin therapy, or at Screening Visit 2 in statin washout subjects.
- 5. Planned change in diet or exercise habits during participation in the double-blind period, or a significant weight change of >5% in the prior 6 months.
- 6. Subjects who have undergone gastric bypass procedures (gastric lap band is acceptable) or ileal resection or plan to undergo either of these procedures.
- 7. History of biliary diversion.
- 8. Uncontrolled diabetes defined as HbA1c ≥9.5% within 60 days prior to randomization (Day 1).
- 9. Administration of any of the following medications as specified below:
  - Prohibited 30 days prior to Day 1:
    - bile acid sequestrants (BAS) including cholestyramine and its derivatives, colesevelam, colestipol, or
    - omega-3 fatty acid containing dietary supplements

- Prohibited <u>3 months</u> prior to Day 1:
  - nicotinic acid and derivatives, ezetimibe, or
  - any prescription or over-the-counter medication or herbal remedy with putative NASH efficacy (except Vitamin E or TZDs), or
  - ursodeoxycholic acid, or
  - fenofibrate or other fibrates, or
  - Any over-the-counter or health foods used to treat lipids including plant sterols and berberine
- Prohibited <u>6 months</u> prior to Day 1:
  - azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate, mofetil, pentoxifylline; budesonide and other systemic corticosteroids; or
  - potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin)
- Prohibited <u>12 months</u> prior to Day 1:
  - antibodies or immunotherapy directed against interleukins, or
  - other cytokines or chemokines
- 10. Evidence of other forms of known chronic liver disease including but not limited to:
  - Positive test result at Screening for hepatitis B surface antigen
  - Active hepatitis C virus (HCV) infection (positive for HCV ribonucleic acid [RNA] at Screening) or history of positive HCV RNA test result
  - PBC, PSC, autoimmune hepatitis or overlap syndrome
  - Alcoholic liver disease
  - Wilson's disease or hemochromatosis or iron overload as defined by presence of 3+ or 4+ stainable iron on liver biopsy
  - Alpha-1-antitrypsin (A1AT) deficiency as defined by diagnostic features in liver histology (confirmed by A1AT level less than normal; exclusion at the Investigator's discretion)
  - Prior known drug-induced liver injury within 5 years before Day 1
  - Known or suspected HCC
- 11. History of liver transplant, current placement on a liver transplant list, or current Model for End-Stage Liver Disease (MELD) score >12. Subjects who are placed on a transplant list despite a relatively early disease stage (eg, per regional guidelines) may be eligible as long as they do not meet any of the other exclusion criteria.

- 12. Presence of hepatic decompensation including:
  - Gastroesophageal varices
  - Ascites
  - Hepatic encephalopathy
  - Spontaneous bacterial peritonitis
  - Hepatorenal or hepatopulmonary syndromes
- 13. Total bilirubin ≥2x upper limit of normal (ULN) at any Screening Visit (subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >2x ULN if their conjugated bilirubin is <2x ULN)
- 14. Creatine phosphokinase (CPK) >5x ULN at Screening Visit 2
- 15. Serum creatinine ≥1.5 mg/dL at any Screening Visit
- 16. Serum ALT >300 U/L at any Screening Visit
- 17. Platelet count <75 000 /mm<sup>3</sup> at any Screening Visit
- 18. Known positivity for human immunodeficiency virus (HIV) infection
- 19. Subjects with recent history (within 1 year of randomization) of cardiovascular disease or with history or planned cardiovascular interventions to treat atherosclerotic cardiovascular disease, including:
  - a) Peripheral or Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting)
  - b) Coronary angioplasty, stenting, or carotid atherectomy
  - c) Cardiac pacemaker or defibrillator (placement of cardiac pacemaker or defibrillator for reasons other than atherosclerotic cardiovascular disease [eg, for treatment of atrial fibrillation subsequent to nodal ablation] is not exclusionary)
  - d) Prosthetic heart valves
  - e) Myocardial infarct, unstable angina, or acute coronary syndrome
  - f) Other clinically significant atherosclerotic cardiovascular disease
  - g) Cerebrovascular accident (stroke), cerebrovascular ischemia, or transient ischemic attack
  - h) Unstable hypertension
  - i) Familial hypercholesterolemia or other genetic lipid abnormality
- 20. Other concomitant disease, malignancy, or condition likely to significantly decrease life expectancy to <5 years, including known cancers (except carcinomas in situ or other stable, relatively benign conditions such as chronic lymphocytic leukemia) and moderate to severe congestive heart failure.
- 21. Known substance abuse, including inhaled or injected drugs in the year before Screening

22. For female subjects: pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the study, or breastfeeding

- 23. Participation in a clinical research study with any investigational product being evaluated for the treatment of diabetes or NASH in the 6 months before Day 1
- 24. Receipt of any investigational product not being evaluated for the treatment of diabetes or NASH from Screening Visit 1 to Day 1, within 30 days prior to Day 1, or within 5 half-lives of the compound before Day 1 (whichever was longer)
- 25. Previous exposure to OCA
- 26. History of known or suspected clinically significant hypersensitivity to OCA or any of its components
- 27. Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain
- 28. Any other condition which, in the opinion of the Investigator, would impede compliance or hinder completion of the study
- 29. Acute cholecystitis or acute biliary obstruction

# 8.4. Subject Withdrawal Criteria

# 8.4.1. Reasons for Mandatory Discontinuation of Investigational Product or Atorvastatin

# 8.4.1.1. Adverse Events ≥Grade 3 in Severity and Possibly, Probably, or Definitely Related to Investigational Product

If a subject experiences an AE that is ≥Grade 3 in severity (Section 12.1.4) that is considered possibly, probably, or definitely related to investigational product, the investigational product must be discontinued.

# 8.4.1.2. Pregnancy

Whenever the site is notified of a possible pregnancy, the subject should be asked to come in for an unscheduled visit to perform a serum pregnancy test. If a female subject becomes pregnant, she must discontinue treatment with investigational product and atorvastatin immediately, but should continue with the study visit schedule and must be followed by the Investigator through pregnancy outcome. The mother (and infant) will be followed as considered appropriate by the Investigator and the Medical Monitor. As described in Section 12.1.8.1, pregnancy is not considered an AE for reporting purposes.

# 8.4.1.3. Severe Drug-Induced Liver Injury

If a subject develops signs and symptoms of a severe drug-induced liver injury, regardless of causality, investigational product and atorvastatin should be interrupted until the event has resolved or returned to baseline, but the subject should continue with the study visit schedule. Subjects who develop significant drug-induced liver injury, which is considered to be causally

related to the investigational product or atorvastatin, should be discontinued from investigational product or atorvastatin, as appropriate and should not be rechallenged. Significant injury as described in Appendix B, and includes evidence of functional hepatic impairment as indicated by rising bilirubin or INR. Natural progression of the underlying condition and other causal factors such as a common bile duct stone or development of other concurrent liver disease should be considered before the investigational product is permanently discontinued.

Severe drug induced-liver injury that is not considered related to investigational product or atorvastatin must be discussed with the Sponsor before investigational product or atorvastatin is reinitiated. Follow-up procedures for subjects resuming treatment, including laboratory evaluations and physical examinations, must be performed after a maximum of 2 weeks of re-treatment and may be conducted at a local clinic if the subject is unable to return to this site. Results must be reported immediately to the site so the Investigator can determine if the subject is to be allowed to continue treatment. Subjects who discontinue due to significant drug-induced liver injury must be followed until the AE has resolved, stabilized, or is not of clinical concern.

#### 8.4.1.4. Myonecrosis

Moderate myonecrosis as defined by creatine kinase  $\geq 10x$  the untreated baseline levels or ULN. Muscle-related symptoms that do not necessitate mandatory discontinuation of investigational product or atorvastatin are detailed in Section 5.8.

## 8.4.2. Reasons for Mandatory Interruption of Investigational Product

# 8.4.2.1. Adverse Events ≥Grade 4 in Severity and Not or Unlikely Related to Investigational Product

If a subject experiences an AE categorized as ≥Grade 4 in severity and not or unlikely related to investigational product, at least a mandatory interruption of investigational product is required.

## 8.4.2.2. Suspected Mild or Moderate Drug-Induced Liver Injury

Because transient fluctuations of ALT or AST are common, and progression to severe drug-induced liver injury or acute liver failure is uncommon, automatic discontinuation of investigational product with an elevation of ALT or AST that is >3x ULN/baseline/nadir or total bilirubin >2x ULN/baseline/nadir, as described in Appendix B, may be unnecessary. If a subject develops signs of a mild or moderate event of drug-induced liver injury, regardless of causality, investigational product should be interrupted until the event has resolved or returned to baseline, but the subject should continue with the study visit schedule. The subject may restart treatment after resolution of the event or return to baseline. Follow-up procedures, including laboratory evaluations and physical examinations, must be performed after a maximum of 2 weeks of re-treatment and may be conducted at a local clinic if the subject is unable to return to the site. Results must be reported immediately to the site so the Investigator can determine if the subject will be allowed to continue treatment.

# 8.4.3. Other Reasons for Study or Treatment Discontinuation of Subjects

A reasonable effort must be made to determine the reason(s) why a subject fails to return for his/her final visit or is discontinued from the study. This information and date must be recorded on the appropriate electronic case report form (eCRF). The following events are considered appropriate reasons for a subject to discontinue from the study:

- The subject decides that it is in his/her best interest. It is fully understood that all subjects volunteer for the study and that they may withdraw their consent to continue in the study at any time
- The Investigator or Sponsor considers that it is advisable or in the best interest of the subject
- There is a major violation of the clinical study protocol
- Noncompliance of the subject
- An inability to provide plasma or urine samples

# 8.4.4. Subject Discontinuation Notification

The Investigator must notify the Sponsor as soon as possible if any subject prematurely discontinues from the study. The date when the subject is withdrawn and the reason for discontinuation must be recorded in the eCRF; additional information may be requested by the Sponsor to complete a discontinuation narrative. Subjects will be considered "lost to follow-up" only after reasonable, documented attempts to reach the subject prove unsuccessful. In all cases, a reasonable effort must be made to determine the reason(s) that a subject fails to return for required study visits or discontinues from the study. This information must be documented in the eCRF.

If a subject is withdrawn from the study early (regardless of the cause), all of the ET evaluations, with the exception of PK procedures, should be performed at the time of withdrawal, to the extent possible.

# 9. TREATMENT OF SUBJECTS

# 9.1. Investigational Product and Atorvastatin Treatment Regimen

While placebo, OCA, and atorvastatin are all study medications provided by the Sponsor, for the purposes of this protocol, investigational product refers to OCA or placebo, and study medication, where used, refers to atorvastatin.

Four treatment groups will be evaluated: placebo, OCA 5 mg, OCA 10 mg, and OCA 25 mg. Each dose will be made up of 1 tablet (ie, 1 placebo tablet, 1 OCA 5-mg tablet, 1 OCA 10-mg tablet, or 1 OCA 25-mg tablet). The list of excipients included in the tablets are provided in the IB.

Investigational product will be taken orally with water, once daily for the duration of the study. Subjects will be instructed to begin dosing on Day 1 and are to take investigational product at

approximately the same time each day. Subjects must be instructed to swallow the tablets whole with water; they must not chew, divide, or crush the tablets.

#### 9.1.1. Double-Blind Period

Subjects enrolled in the study will be randomized to receive one of the following treatments: OCA 5 mg, OCA 10 mg, OCA 25 mg, or placebo, starting on Day 1.

At the Week 4 Visit, all subjects will also initiate treatment with atorvastatin at a dose of 10 mg once daily. At the Week 8 Visit, atorvastatin will be increased to 20 mg once daily (if 10 mg daily is tolerated), and continued for an additional 4 weeks. After 4 weeks of treatment at 20 mg, the atorvastatin dose may be titrated (up or down) at the Week 12 Visit as clinically indicated using the atorvastatin prescribing information and the guidance for lipid management (see Appendix A). Blinded treatment with investigational product and open-label atorvastatin will continue through the Week 16 Visit. Investigational product will be dispensed in bottles of 30 tablets

#### 9.1.2. LTSE

Subjects who complete the Week 16 Visit of the double-blind phase will be able to participate in an open-label LTSE. The Week 16 Visit of the double-blind phase will be Day 1 of the LTSE phase of the study.

Following completion of Week 16 Visit procedures, all subjects will be treated with open-label OCA 10 mg or OCA 25 mg. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will be randomized in a 1:1 ratio to receive OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg or OCA 25 mg during the double-blind phase will continue on the same dose throughout the LTSE.

Investigational product during the LTSE period will be dispensed in bottles of 30 or 100 tablets, and subjects will be instructed to take one or more tablets per day per his/her OCA dose assignment. During the LTSE phase, the dose of atorvastatin may remain the same as during the double-blind phase or may be modified as clinically indicated per atorvastatin prescribing information and lipid management guidelines (Appendix A).

#### 9.2. Concomitant Medications

Relevant information about all concomitant medications (including prescribed, over-the-counter, or herbal preparations) taken prior to (ie, within 12 months of Day 1) and during the study must be recorded in the source documents and eCRF, as well as any dose or dose regimen changes that occur during the study.

# 9.2.1. Medications with Potential NASH-Modifying Properties

Doses of TZDs and Vitamin E should be stable 6 months before Day 1 through Week 16. Ideally, subjects should generally remain on baseline TZDs and/or Vitamin E throughout both the double-blind and LTSE phases of the study unless the baseline therapy is no longer considered clinically appropriate by the Investigator.

# 9.2.2. Diabetes-Specific Therapy

All diabetes-specific therapies except TZDs should be at a stable dose for ≥3 months prior to Day 1 through Week 16. TZDs must be at a stable dose for ≥6 months prior to Day 1 through Week 16. Ideally, subjects should remain on Baseline diabetes-specific therapies through the end of the LTSE, but will be allowed to make changes if the Baseline therapy is no longer considered clinically appropriate by the Investigator.

#### 9.2.3. Management of Changes in Cholesterol

During the double-blind phase of the study, the dose of atorvastatin administration should be as described in this protocol through Week 12 unless tolerability issues develop as referenced in Section 7.4.2. At the Week 12 Visit, Investigators may increase or decrease the dose of atorvastatin as clinically indicated.

During the LTSE, Investigators may add or change the management of treatment as clinically appropriate. Appendix A provides a general guidance for cholesterol management including monitoring, triggers for intervention, and treatment goals.

#### 9.2.4. Prohibited Medications

The medications prohibited per the study enrollment exclusion criteria and or during the study are listed below and summarized in Table 3:

- Prohibited <u>30 days</u> prior to Day 1:
  - BAS including cholestyramine, colesevelam, colestipol, or
  - omega-3 fatty acid containing dietary supplements
- Prohibited 3 months prior to Day 1 and throughout the double-blind period:
  - nicotinic acid and derivatives, ezetimibe, or
  - fenofibrate or other fibrates
  - any over-the-counter or health foods used to treat lipids including plant sterols and berberine
- Prohibited 3 months prior to Day 1 and throughout the double-blind period and LTSE:
  - any prescription or over-the-counter medication or herbal remedy with putative NASH efficacy (except Vitamin E or TZDs)
  - ursodeoxycholic acid
- Prohibited 6 months prior to Day 1 and throughout the double-blind period and LTSE:
  - azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate, mofetil, pentoxifylline; budesonide and other systemic corticosteroids;

potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin)

- Prohibited 12 months prior to Day 1 and throughout the double-blind period:
  - antibodies or immunotherapy directed against interleukins or
  - other cytokines or chemokines
- Prohibited throughout the double-blind phase of the study:
  - weight loss drugs including appetite suppressants (eg, orlistat, lorcaserin)
  - medications contraindicated in the atorvastatin label, including HIV and Hepatitis C protease inhibitors, clarithromycin, and itraconazole (refer to atorvastatin prescribing information in Appendix E for complete list). These medications are also prohibited during the LTSE phase if the subject continues to receive atorvastatin during the LTSE.
- Prohibited during the double-blind and LTSE phases of the study:
  - medications historically associated with NAFLD including: amiodarone, tetracyclines, tamoxifen, estrogens (at doses greater than those used for hormone replacement), anabolic steroids

Table 3: Medications Prohibited Prior to Randomization and/or During Study Participation

| | Use | e Prohibited Pric | Use Prohibited During Study | | | |
|---|---|---|---|---|---|---|
| Medications | -12 Months | -6 Months | -3 Months | -30 Days | Double-Blind<br>Phase | LTSE |
| Bile acid sequestrants including cholestyramine, colesevelam, colestipol | | | | X | | |
| Omega-3 fatty acid containing dietary supplements | | | | X | | |
| Nicotinic acid and derivatives | | | X | X | X | |
| Ezetimibe | | | X | X | X | |
| Fenofibrate or other fibrates | | | X | X | X | |
| Any over-the-counter or health foods used to treat lipids including plant sterols and berberine | | | X | X | X | |
| Any prescription or over-the-counter medication or herbal remedy with putative NASH efficacy (except Vitamin E or TZDs ) | | | X | X | X | X |
| Ursodeoxycholic acid | | | X | X | X | X |
| Azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate, mofetil, pentoxifylline; budesonide and other systemic corticosteroids | | X | X | X | X | X |
| Potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin) | | X | X | X | X | X |

**Table 3:** Medications Prohibited Prior to Randomization and/or During Study Participation (Continued)

| | Use | e Prohibited Pric | Use Prohibited During Study | | | |
|---|---|---|---|---|---|---|
| Medications | -12 Months | -6 Months | -3 Months | -30 Days | Double-Blind<br>Phase | LTSE |
| Antibodies or immunotherapy directed against interleukins | X | X | X | X | X | |
| Other cytokines or chemokines | X | X | X | X | X | |
| Weight loss drugs including appetite suppressants (eg, orlistat, lorcaserin) | | | | | X | |
| HIV and Hepatitis C protease inhibitors, clarithromycin, itraconazole | | | | | X | X |
| Medications historically associated with NAFLD including: amiodarone, tetracyclines, tamoxifen, estrogens (at doses greater than those used for hormone replacement), anabolic steroids | | | | | X | X |

Note: For clarity, only prior months and study periods with prohibited use are indicated with "X"; other periods with no restrictions are shaded grey.

#### 9.2.5. Standard of Care and Other Concomitant Medications

With the exception of Vitamin E, TZDs and other diabetes-specific therapy, allowed concomitant medications should be at a stable dose 30 days before Day 1. Concomitant medications will be used at the discretion of the usual care provider (or Investigator if also the usual care provider). Relevant information about all concomitant medications taken before (ie, within 12 months of Day 1; Table 3) and during the study must be recorded in the source documents and eCRF, as well as any dose or dose regimen changes that occur during the study.

Subjects taking BAS (including cholestyramine and its derivatives, colestipol, colesevelam, or other sequestrants) or aluminum hydroxide- or smectite-containing antacids should be instructed to stagger their dosing of investigational product, ensuring at least 4 hours between doses of the BAS and/or antacids and the investigational product (ie, BAS should be administered 4 hours before or 4 hours after investigational product administration).

Taken concomitantly, OCA and warfarin may decrease INR, thus INR should be monitored and the dosage of warfarin adjusted, as needed, to maintain the target INR range.

The effect of OCA on drug metabolizing enzymes has been evaluated in both in vitro and clinical studies. The PK profile of caffeine, a sensitive CYP1A2 substrate, showed weak effect of OCA on CYP1A2. Based on these results, OCA may increase the exposure of narrow therapeutic index drugs that are substrates for CYP1A2, such as theophylline and tizanidine.

# **9.3.** Treatment Compliance

The Investigator should assess the subject's compliance with dosing of investigational product and open-label atorvastatin on an ongoing basis throughout the study and confirm by conducting drug accountability (ie, count of returned tablets) during subjects' onsite visits.

Subjects should be instructed to retain all bottles of investigational product and atorvastatin, even if empty, and to return them to the Investigator at the subsequent visit (refer to Table 1 and Table 2). The Investigator or designee should perform drug accountability and, if applicable, follow up with the subject to retrieve any investigational product and atorvastatin bottles that have not been returned.

If the Investigator has concerns about a subject's dosing compliance s/he should discuss this with the subject, assess the reasons for noncompliance and the likelihood that the subject will remain noncompliant, and notify the Sponsor accordingly. Continued study eligibility should be assessed based on the subject's compliance with investigational product and atorvastatin dosing and clinic visits.

# 9.4. Randomization and Blinding

The initial phase of the study will be conducted in a double-blind, placebo-controlled manner. Enrolled subjects will be randomized in a 1:1:1:1 ratio to 1 of 4 treatment groups (OCA 5 mg, OCA 10 mg, OCA 25 mg, or placebo) based on a predefined randomization code (generated by Sponsor or designee) using an IWRS. The IWRS will serve as the investigational product inventory and management system and may be integrated with the study database.

The Investigator or designee will be required to register the subject in the IWRS and may be prompted to provide patient data necessary to properly randomize and allocate the subject to treatment. A randomization number will be assigned and investigational product (OCA or placebo) dispensing information will be provided (eg, bottle numbers allocated) while maintaining the study blind. The subjects, Investigator, and study site staff will be blinded to the subjects' treatment allocation in the double-blind phase of the study until all subjects have completed the double-blind phase of the study and the database is locked.

In the LTSE phase, all subjects will be treated with open-label OCA 10 mg or OCA 25 mg: subjects randomized to placebo or OCA 5 mg during the double-blind phase will be randomized in a 1:1 ratio to receive OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase, and subjects randomized to OCA 10 mg or OCA 25 mg during the double-blind phase will continue on the same dose throughout the LTSE.

#### 9.4.1. Stratification

In order to ensure that factors with the potential to affect treatment response are randomized in equal proportions to the different treatment groups, subjects will be stratified by LDL cholesterol concentration (Screening Visit 2 LDL cholesterol value for statin washout subjects or Screening LDL cholesterol value for statin-free subjects). Randomization will be stratified by the pre-randomization fasted serum LDL cholesterol concentration (≤125 mg/dl or >125 mg/dL) and baseline fibrosis stage (stage 1, 2 or stage 3, 4).

## 9.4.2. Emergency Unblinding Procedures

Randomization codes and corresponding treatment assignments will be made available to the Investigator and the Medical Monitor for emergency use only through the IWRS system. When possible, the Medical Monitor should be consulted in the event that a medical emergency necessitates unblinding (ie, in situations where knowledge of the blinded treatment is necessary for further medical management of the subject). If it is not reasonable to inform the Medical Monitor in advance of unblinding, the Investigator must promptly document the case in the subject's source record. Subsequently, the Investigator should contact the Medical Monitor to explain any premature unblinding of treatment assignment (eg, accidental unblinding or unblinding due to a serious AE [SAE]). Procedures for unblinding a subject's treatment will be provided separately to the Investigator. The Medical Monitor will document within study correspondence the rationale, circumstances, and the person(s) being informed about the unblinding.

The DMC (refer to Section 13.8) will have access to the IWRS and will be able to unblind individual subjects. The DMC will review aggregate data during closed sessions. The DMC will document details about any subject who was unblinded in the closed session DMC minutes, which will be made available to the Sponsor only after the double-blind database is locked and unblinded.

Access to randomization codes and corresponding treatment assignments will also be made available through the IWRS system to the appropriate, named individual(s) responsible for reporting SAEs and suspected unexpected serious adverse reactions (SUSARs) to the regulatory authorities.

# 9.5. Assignment of Site and Subject Numbers

#### 9.5.1. Site Numbers

Each study site selected to participate in this study will be assigned a Site Number by the Sponsor. The Site Number will be used to categorize subject data and to identify the site and or Investigator within study documents. This number will be recorded in the eCRF.

## 9.5.2. Subject Numbers

Subjects will be identified by a unique 6-digit number. The first 3 digits will represent the site number and the last 3 digits, the Screening number, which will be assigned sequentially by the site

#### 9.6. Restrictions

# 9.6.1. Fasting Requirement at Study Visits

All subjects must have been fasting for at least 8 hours prior to Screening Visit 2 (Week -1 Visit) and all subsequent study visits, as all analytes will be assayed in fasting blood, serum, or plasma samples (Table 1 and Table 2). Water is permitted during the fasting period.

If the subject reports having eaten within 8 hours, the information will be documented accordingly in the source and eCRF and the subject will be reminded that at least 8-hour fasting is required prior to all study visits, but water is permitted. The blood sample will still be collected during the visit with the exception of Screening Visit 2, which will require rescheduling of the visit.

## 9.6.2. Grapefruit and Grapefruit Juice

Grapefruit and grapefruit juice consumption should be discouraged following initiation of atorvastatin due to possible increases in plasma concentration of atorvastatin (please refer to atorvastatin prescribing information [Appendix E]).

#### 9.6.3. Diet and Exercise

Consistent with the exclusion criteria (Section 8.3), subjects should not make significant changes to their diet and exercise habits during the double-blind phase. This is not intended to override physician advice for lifestyle modification, and inclusion in the study should preferably be after lifestyle modifications have been made and are stable.

### 9.7. Visit Procedures

## 9.7.1. Visit Windows

All Screening assessments should occur  $\leq$ 35 days prior to the Randomization/Day 1 Visit. Subjects who are taking statins at the time of screening or within 30 days of Screening Visit 1 are required to stop statin therapy for 4 weeks (28 ( $\pm$ 1) days), and provide a fasting blood sample at Screening Visit 2 to confirm eligibility. Subjects who have not taken statins within 30 days of Screening Visit 1 are not required to enter into the washout period and may proceed to Screening

Visit 2 to provide a fasting blood sample. The Randomization/Day 1 Visit may occur as soon as all screening labs are available and eligibility is confirmed.

All visits during the double-blind phase will be relative to Day 1 (eg, if the Week 2 Visit occurs 4 days late, the Week 4 Visit should still be 4 weeks from Day 1), and should occur within ±4 days of the visit day. The timing of all study visits during the LTSE is relative to Week 16/LTSE Day 1. LTSE Visits should occur within ±1 week of the visit day.

The visit windows are summarized below:

| Visit or Procedure | Visit Window and/or Interval |
|---|---|
| Screening Visit 1 | Visit(s) are to occur ≤5 weeks (35 days) prior to Day 1. |
| Screening Visit 2 (Week -1) | ±1 day |
| Randomization (Day 1) | This is the day of Randomization and the first day of dosing with investigational product. On-treatment visit scheduling should be calculated from this point going forward unless stated otherwise. |
| Week 2, Week 4, Week 8, and<br>Week 12 | ±4 days; the visits during double-blind phase will be relative to Day 1 (ie, first dose of investigational product) |
| Week 6, Week 10, and Week 14 (Contact visits) | ±4 days |
| Week 16 (LTSE Day 1) | ±4 days |
| LTSE Visits: Month 1, Month 3,<br>Month 6, Month 9, Month 12,<br>Month 15, Month 18, and Month 21 | ±1 week (7 days); the LTSE visits are relative to LTSE Day 1 (ie, Week 16 of double-blind phase) |
| EOS | ±1 week (7 days) relative to the EOS date announced by the Sponsor |
| ET | As soon as possible upon study discontinuation and as near as possible to last dose taken |

EOS = End of Study; ET = Early Termination

#### 9.7.2. Informed Consent Procedures

The Investigator or designee will explain the nature, purpose possible risks and benefits of the study to the subject and will provide him/her with a copy of the written information and informed consent form (ICF). The subject will be given sufficient time to consider the study before deciding whether or not to participate. The subject will be informed that participation is voluntary and that his/her future medical treatment will not be compromised by participation in the study and that he or she can withdraw from the study at any time. The subject must be willing and able to provide written informed consent before entering the study. The Investigator or a medically qualified designee is responsible for administering and documenting the written informed consent of the subject. The subject will be given a copy of the written information sheet and his/her signed and dated consent form). At selected study sites, subjects will have the option to consent to participate in an additional PK assessment. Subjects may also be required to sign a new consent form prior to entering the LTSE phase of the study. Subjects will be requested to provide blood samples for exploratory future analysis of analytes such as adiponectin, plasminogen activator inhibitor-1(PAI-1), and B-type natriuretic peptide (BNP; Table 10).

## 9.7.3. Screening Visit 1 Procedures

The Screening Visit assessments must be performed  $\leq$ 5 weeks prior to Day 1 to determine whether the subject meets all the inclusion criteria and none of the exclusion criteria. Subjects who do not fulfill all eligibility criteria will not be enrolled in the study.

Subjects who are statin-free (ie, no statin use within 30 days of Screening) must return for fasted serum chemistry labs at Screening Visit 2, and may proceed to the Randomization/Day 1 Visit once screening labs are available and eligibility is confirmed; subjects who need to wash out statin therapy are required to return for Screening Visit 2 following the washout period.

Screening Visit procedures for all subjects are as follows:

- Review ICFs and obtain signatures before performing any study-related procedures, including Screening procedures.
- Collect medical history.
- Verify inclusion and exclusion criteria for eligibility.
- Perform a physical examination.
- Perform a standard 12-lead electrocardiogram (ECG).
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference, and height.
- Determine alcohol consumption (using AUDIT questionnaire).
- Assess availability of liver biopsy samples: If >1 year since last biopsy, schedule pretreatment biopsy. Liver biopsies conducted within 1 year of Day 1, for which unstained slides can be obtained and submitted for central review, are considered adequate for study entry. All samples must be submitted for central read such that the report is available prior to Day 1.
- For participating sites only: TE is scheduled for Screening Visit 1; however, it may be performed any time between Screening Visit 1 and prior to Randomization (Day 1). In addition, if TE has been done within 3 months of Day 1 and a report/adequate data is/are available, a pretreatment TE at Day 1 is not required.
- Assess and record any pretreatment-emergent AEs (after the ICF has been signed).
- Record prior (if within 12 months of Day 1) and current concomitant medications.
- Obtain serum sample for hepatitis B surface antigen or hepatitis C antibody (and positive HCV ribonucleic acid [RNA]) testing to confirm study eligibility.
- Schedule laboratory visit for fasted blood samples for
  - Serum chemistry (includes basic lipid panel and liver biochemistry panel), hematology, and coagulation

- Obtain urine sample for urinalysis.
- Perform serum pregnancy test in females of childbearing potential.
- Instruct the subject to fast overnight (at least 8 hours) before the next visit (water is permitted).

Additional Screening Visit 1 procedure for subjects currently taking statins:

• Subjects who are currently taking statins, defined as statin use within 30 days of Screening, will be instructed to discontinue statin therapy following Screening Visit 1. After 4 weeks of statin washout, subjects will return for Screening Visit 2 to provide blood samples for fasted serum chemistry.

## 9.7.4. Screening Visit 2 Visit Procedures

All subjects will return for Screening Visit 2 to confirm eligibility criteria and provide blood samples for fasted serum chemistry.

For subjects who were receiving statin therapy at the time of screening:

• Verify that subjects have completed a 4-week washout period.

## For all subjects:

- Review inclusion and exclusion criteria for eligibility.
- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, the visit should be rescheduled.
- Obtain blood samples for
  - Serum chemistry (will include basic lipid and liver biochemistry panel), hematology, and coagulation
  - CPK
- Assess and record pretreatment-emergent AEs.
- Assess and record new concomitant medications.
- For participating sites only: Perform TE if not done during Screening Visit 1 or a report/adequate data from a scan done within 3 months and Day 1 is/are not available.

## 9.7.5. Randomization/Day 1 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that at least 8-hour fasting is required prior to all study visits, but water is permitted.

- Review inclusion and exclusion criteria for eligibility.
- Perform a standard 12-lead ECG.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, and waist and hip circumference.
- Determine alcohol consumption (using AUDIT questionnaire).
- Assess and record any pretreatment-emergent AEs.
- Record prior (since Screening Visit 1) and current concomitant medications.
- For participating sites only: Perform TE if not done during Screening Visit 1 or Screening Visit 2, or if a report/adequate data from a scan done within 3 months and Day 1 is/are not available.
- Obtain blood samples for:
  - Serum chemistry (includes basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - CPK, if myopathy suspected
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - Blood sample for future exploratory analysis of biomarkers adiponectin, PAI-1, and BNP
  - Thyroid Function Tests: TSH, T4, and T3
  - Possible analysis of conjugated and unconjugated bile acids
- Obtain urine sample for urinalysis.
- Perform a urine-based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Randomize the subject only if s/he meets all inclusion criteria and no exclusion criteria: Record the visit in IWRS along with the subject's Screening Visit 2 (Week -1) fasting LDL cholesterol value, randomize the subject to study treatment group, and dispense investigational product according to IWRS instructions.
- Administer the first dose of investigational product at the study site. Instruct the subject to swallow the tablet whole with water; s/he must not chew, divide, or crush the tablet.

- Schedule the next visit, reiterate dosing instructions, and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product on the morning of the next visit
  - To bring the investigational product bottle(s); s/he will dose at the clinic
  - To fast overnight (at least 8 hours) before the next visit, but water is permitted

# Additional Day 1 Procedures for PK Subjects

At participating investigational sites, subjects will have the option to consent to participate in an additional PK assessment. This is optional and subjects may decline to participate without affecting their involvement in the rest of the study.

Following collection of the Day 1 fasted samples indicated above, subjects who are participating in the PK assessment will each receive a single dose of their assigned investigational product with water. Serial blood samples will be obtained for measurement of OCA and its conjugates 30 minutes prior to dosing and at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until the 1-hour sample is collected. Meal will be provided following collection of the 1-hour PK sample, and will be a meal replacement drink with nutrition information that has been submitted to and approved by the Sponsor in advance.

## 9.7.6. Week 2 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference.
- Assess and record AEs.
- Review and record concomitant medications.
- Collect used bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.
- Obtain blood samples for:
  - Serum chemistry (includes basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes

- CPK, if myopathy suspected
- Perform a urine-based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Schedule the next visit, reiterate dosing instructions and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product on the morning of the next visit
  - To bring the investigational product bottle(s); s/he will dose at the clinic
  - To fast overnight (at least 8 hours) prior to the next visit, but water is permitted

#### 9.7.7. Week 4 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference.
- Assess and record AEs.
- Review and record concomitant medications.
- Collect used bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.
- Obtain blood samples for:
  - Serum chemistry (includes basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected
- Perform a urine-based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.

 Record the visit in IWRS and dispense investigational product and atorvastatin as instructed.

- Administer the daily dose of investigational product at the study site. Instruct the subject to swallow the tablet whole; s/he must not chew, divide, or crush the tablet.
- Administer the daily dose of atorvastatin at the study site. Instruct the subject to swallow the tablet whole; s/he must not chew, divide, or crush the tablet.
- Schedule the next visit, reiterate dosing instructions and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product or atorvastatin on the morning of the next visit
  - To bring the investigational product and atorvastatin bottle(s); s/he will dose at the clinic
  - To fast overnight (at least 8 hours) prior to the next visit. Fasting is required prior to all study visits, but water is permitted.

# 9.7.8. Week 6 Safety Contact

- This is a telephone contact with the subject to
  - Review and record AEs
  - Review and record concomitant medications
  - Assess investigational product and atorvastatin compliance

#### 9.7.9. Week 8 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference
- Assess and record AEs.
- Review and record concomitant medications.
- Collect used bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.

• Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability.

- Obtain blood samples for:
  - Serum chemistry (includes basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected
  - Blood sample for future exploratory analysis of biomarkers adiponectin, PAI-1, and BNP
- Perform a urine-based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Record the visit in IWRS and dispense investigational product and atorvastatin as instructed.
- Administer the daily dose of investigational product at the study site. Instruct the subject to swallow the tablet whole; s/he must not chew, divide, or crush the tablet.
- Administer the daily dose of atorvastatin at the study site. Instruct the subject to swallow the tablet whole; s/he must not chew, divide, or crush the tablet.
- Reiterate dosing instructions and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product or atorvastatin on the morning of the next visit
  - To bring the investigational product and atorvastatin bottle(s); s/he will dose at the clinic
  - To fast overnight (at least 8 hours) prior to the next visit. Fasting is required prior to all study visits, but water is permitted.

## 9.7.10. Week 10 Safety Contact

- This is a telephone contact with the subject to:
  - Review and record AEs
  - Review and record concomitant medications
  - Assess investigational product and atorvastatin compliance

#### 9.7.11. Week 12 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference.
- Assess and record AEs.
- Review and record concomitant medications.
- Collect used bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.
- Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability.
- Obtain blood samples for:
  - Serum chemistry (includes basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected
- Perform a urine-based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Record the visit in IWRS and dispense investigational product and atorvastatin as instructed.
- Administer the daily dose of investigational product at the study site. Instruct the subject to swallow the tablet whole; s/he must not chew, divide, or crush the tablet.
- Administer the daily dose of atorvastatin at the study site. Instruct the subject to swallow the tablet whole; s/he must not chew, divide, or crush the tablet.
- Reiterate dosing instructions and advise the subject:
  - Take the investigational product at approximately the same time each day

 NOT to take investigational product or atorvastatin on the morning of the next visit

- To bring the investigational product and atorvastatin bottle(s); s/he will dose at the clinic
- To fast overnight (at least 8 hours) prior to the next visit. Fasting is required prior to all study visits; water is permitted.

# 9.7.12. Week 14 Safety Contact

- This is a telephone contact with the subject to:
  - Review and record AEs
  - Review and record concomitant medications
  - Assess investigational product and atorvastatin compliance

#### 9.7.13. Week 16 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Perform a physical examination.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference.
- Perform a standard 12-lead ECG.
- Determine alcohol consumption (using AUDIT questionnaire).
- For participating sites only: perform TE
- Assess and record AEs.
- Review and record concomitant medications.
- Collect all used and unused bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.
- Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability.
- Obtain blood samples for:
  - Serum chemistry (includes basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected
  - Blood sample for future exploratory analysis of biomarkers adiponectin, PAI-1, and BNP
  - Thyroid Function Tests: TSH, T4, and T3
  - Possible analysis of conjugated and unconjugated bile acids
- Obtain urine sample for urinalysis.
- Perform a urine-based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Record the visit in IWRS and indicate if the subject is continuing into the LTSE.

#### 9.7.13.1. Additional Week 16 Procedures for PK Subjects

At participating investigational sites, subjects will have the option to consent to participate in an additional PK assessment. This is optional and subjects may decline to participate without affecting their involvement in the rest of the study. Consent to participate in the assessment can be given at any point during study participation prior to the Week 16 Visit.

Following collection of the Week 16 fasted samples indicated above, subjects who are participating in the PK assessment will each receive a single dose of their assigned double-blind investigational product with water. Serial blood samples will be obtained for measurement of OCA and its conjugates, and atorvastatin and its metabolites, 30 minutes prior to dosing and at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until the 1-hour sample is collected. The meal will be provided following collection of the 1-hour PK sample, and will be a meal replacement drink with nutrition information that has been submitted to and approved by the Sponsor in advance.

# 9.7.14. Additional Procedures at Week 16/LTSE Day 1 Visit for Subjects Continuing into the LTSE

Subjects who continue into the LTSE phase after completing the procedures listed for the Week 16 Visit (Section 9.7.13) will undergo the following procedures after signing the LTSE-specific ICF:

 Record the visit in IWRS, randomize the subject to one of the open-label treatment groups, and dispense open-label investigational product according to IWRS instructions.

- If the subject is continuing with atorvastatin therapy, dispense (via IWRS) and provide dosing instructions as clinically indicated (Appendix A).
- Reiterate dosing instructions for investigational product and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product or atorvastatin on the morning of the next visit
  - To bring the investigational product and atorvastatin bottle(s); s/he will dose at the clinic
  - To fast overnight (at least 8 hours) prior to the next visit. Fasting is required prior to all study visits, but water is permitted.

#### 9.7.15. Early Termination/End of Study Procedures: Double-Blind Period

Subjects who terminate participation in the study prior to the Week 16 Visit should have an early termination (ET) Visit as soon as possible following the decision to discontinue therapy. If the study is terminated early by the Sponsor (Section 7.5), the subject will be asked to return to the site for ET/EOS procedures as soon as possible. The procedures to be performed at the double-blind phase ET/EOS Visit are as follows:

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Perform a physical examination.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference.
- Perform a standard 12-lead ECG.
- Determine alcohol consumption (using AUDIT questionnaire).
- For participating sites only: perform TE
- Assess and record AEs.
- Review and record concomitant medications.

• Collect used and unused bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.

- Collect used and unused bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability.
- Obtain blood samples for:
  - Serum chemistry (will include basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected
  - Blood sample for future exploratory analysis of biomarkers adiponectin, PAI-1, and BNP
  - Thyroid Function Tests: TSH, T4, and T3
  - Possible analysis of conjugated and unconjugated bile acids
- Obtain urine sample for urinalysis.
- Perform a urine-based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Obtain urine sample for urinalysis.
- Record the visit in the IWRS.

#### **9.7.16.** LTSE Visits

LTSE Visits should occur within ±1 week of the visit day and the timing of all visits should be relative to the double-blind Week 16 Visit (ie, the start of the LTSE; LTSE Day 1). For example, if the Month 6 Visit occurred 1 week late, the Month 9 Visit should still be approximately 9 months after the Week 16 Visit.

The first LTSE visit following LTSE Day 1 will occur at LTSE Month 1. The next visit will occur at LTSE Month 3 and every 3 months thereafter (eg, at Months 6, 9, and 12) for the duration of the LTSE. The quarterly visit procedures described below will repeat annually for the duration of the LTSE. For example, once a subject completes a year (Month 12 Visit) in the LTSE, their next visit should be 3 months later and the procedures described for the Month 3 LTSE Visit should be followed.

#### 9.7.17. LTSE Month 1 Visit Procedures

• Verify that the subject has fasted for at least 8 hours.

- Record fasting status in the source and eCRF.
- If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record AEs.
- Review and record concomitant medications.
- Collect used bottles of investigational product, assess investigational product compliance, and perform investigational product accountability. Following product accountability, redispense the same bottle of investigational product for use until the next visit.
- Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability. Following atorvastatin accountability, if the subject is continuing with the same dose of atorvastatin, redispense the same bottle for use until the next visit.
  - NOTE: If atorvastatin dose is up-titrated or re-initiated after dose interruption, a
    telephone safety contact must be conducted 2 weeks following the change in dose
    to assess for AEs, concomitant medications, and investigational product and
    atorvastatin compliance.
- Obtain blood samples for:
  - Serum chemistry (will include basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Markers of glucose metabolism
  - CPK, if myopathy suspected
- Perform a urine based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Reiterate dosing instructions for investigational product and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product or atorvastatin (if applicable) or on the morning of the next visit
  - To bring the investigational product and atorvastatin (if applicable) bottle(s); s/he will dose at the clinic
  - To fast overnight (at least 8 hours) prior to the next visit. Fasting is required prior to all study visits, but water is permitted.

## 9.7.18. LTSE Month 3, Month 6, Month 9, Month 15, Month 18, and Month 21 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Perform a physical examination (only at Month 3 and Month 15 Visits).
- Perform a standard 12-lead ECG.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference.
- Determine alcohol consumption (using AUDIT questionnaire [only at Month 6 and Month 18 Visits]).
- Assess and record AEs.
- Review and record concomitant medications.
- Collect used bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.
- Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability.
  - NOTE: If atorvastatin dose is up-titrated or re-initiated after dose interruption, a
    telephone safety contact must be conducted 2 weeks following the change in dose
    to assess for AEs, concomitant medications, and investigational product and
    atorvastatin compliance.
- Obtain blood samples for:
  - Serum chemistry (will include basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses
  - Reverse cholesterol transport analytes (only at Month 6 and Month 18)
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected

 Perform a urine based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.

- Record the visit in IWRS and dispense investigational product and atorvastatin (if applicable) as instructed.
- Reiterate dosing instructions for investigational product and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product or atorvastatin (if applicable) or on the morning of the next visit
  - To bring the investigational product and atorvastatin (if applicable) bottle(s); s/he will dose at the clinic
  - To fast overnight (at least 8 hours) prior to the next visit. Fasting is required prior to all study visits, but water is permitted.

#### 9.7.19. LTSE Month 12 Visit Procedures

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.
  - If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.
- Perform a physical examination.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference
- Perform a standard 12-lead ECG.
- Determine alcohol consumption (using AUDIT questionnaire).
- Assess and record AEs.
- Review and record concomitant medications.
- For participating sites only: Perform TE
- Collect used bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.
- Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability.

- Obtain blood samples for:
  - Serum chemistry (will include basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected
  - Blood sample for future exploratory analysis of biomarkers adiponectin, PAI-1, and BNP
  - Thyroid Function Tests: TSH, T4, and T3
- Obtain urine sample for urinalysis.
- Perform a urine based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Record the visit in IWRS and dispense investigational product and atorvastatin (if applicable) as instructed.
- Reiterate dosing instructions for investigational product and advise the subject:
  - Take the investigational product at approximately the same time each day
  - NOT to take investigational product or on the morning of the next visit, and
  - To bring the investigational product and atorvastatin (if applicable) bottle(s); s/he will dose at the clinic, and
  - To fast overnight (at least 8 hours) prior to the next visit. Fasting is required prior to all study visits, but water is permitted.

#### 9.7.20. LTSE End of Study/Early Termination Procedures

When the LTSE concludes, subjects will be asked to return to the site for EOS procedures as soon as possible. Subjects who terminate participation in the study during the LTSE should have an ET Visit as soon as possible following the decision to discontinue therapy. If the study is terminated by the Sponsor (Section 7.5), the subjects will be asked to return to the site for the ET/EOS procedures as soon as possible. The procedures to be performed at the LTSE ET/EOS Visit are as follows

- Verify that the subject has fasted for at least 8 hours.
  - Record fasting status in the source and eCRF.

 If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is required prior to all study visits, but water is permitted.

- Perform a physical examination.
- Assess and record vital signs (body temperature, sitting heart rate, respiratory rate, and sitting blood pressure).
- Assess and record anthropometric measures: body weight, waist and hip circumference.
- Perform a standard 12-lead ECG.
- Determine alcohol consumption (using AUDIT questionnaire).
- Assess and record AEs.
- Review and record concomitant medications.
- For participating sites only: Perform TE
- Collect used and unused bottles of investigational product, assess investigational product compliance, and perform investigational product accountability.
- Collect used and unused bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability.
- Obtain blood samples for:
  - Serum chemistry (will include basic lipid panel and liver biochemistry panel), hematology, and coagulation
  - Lipoprotein analyses and reverse cholesterol transport analytes
  - PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 10)
  - Vitamin D
  - CPK, if myopathy suspected
  - Blood sample for future exploratory analysis of biomarkers adiponectin, PAI-1, and BNP
  - Thyroid Function Tests: TSH, T4, and T3
- Obtain urine sample for urinalysis.
- Perform a urine based β-hCG pregnancy test in female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential if urine β-hCG pregnancy test is positive.
- Record the visit in IWRS.

#### 9.7.21. Unscheduled Safety Visits

The Investigator may schedule an at-clinic Unscheduled/Safety Visit at any time if clinically warranted or requested by the Medical Monitor. Unscheduled and/or repeat assessments, including additional laboratory tests or investigations, may be conducted.

An increase in aminotransferases (ALT or AST) to >3× baseline (and >ULN) or total bilirubin >2× baseline (and >ULN) should be followed by repeat testing within 48 to 72 hours of the serum chemistry to confirm the abnormalities and to determine if they are increasing or decreasing (Appendix B). AE information should also be collected. If symptoms persist or repeat testing shows ALT >3× baseline (and >ULN) or total bilirubin >2× baseline (and >ULN), subjects should be followed until resolution of the abnormality and as clinically indicated depending on other laboratory and clinical signs and symptoms.

As appropriate, the Medical Monitor should be contacted.

#### 10. INVESTIGATIONAL PRODUCT AND STUDY MEDICATION

#### **10.1.** Investigational Product (OCA or Placebo)

#### **Double-Blind Phase:**

Investigational Product will be supplied as white, round, film-coated tablets containing OCA 5 mg, OCA 10 mg, OCA 25 mg, or placebo. All tablets will be debossed with "INT" on one side and "3547" on the other side, and will be of the same size and appearance. The tablets contain the following inactive ingredients: microcrystalline cellulose, sodium starch glycolate, and magnesium stearate. The 25-mg tablet also contains silicon dioxide. The investigational product tablets will be provided in high-density polyethylene (HDPE) bottles with an induction seal and child-resistant caps. All investigational product will be manufactured according to Good Manufacturing Practice (GMP).

#### LTSE Phase:

10-mg and 25-mg OCA tablets for the LTSE Phase will be supplied as white tablets.

• White OCA tablets are round and debossed with "INT" on one side and "3547" on the other side.

The tablets contain the following inactive ingredients: microcrystalline cellulose, sodium starch glycolate, and magnesium stearate. The 25-mg tablet also contains silicon dioxide. All investigational product will be provided as a tablet for oral administration and provided in HDPE bottles with an induction seal and child-resistant caps.

## 10.2. Investigational Product Packaging and Labeling

The packaging and labeling of investigational product supplies will be performed according to GMP standards by designated, qualified vendors. A designated vendor will also be responsible for the distribution of the investigational product and placebo to the clinical sites.

For the double-blind period, investigational product will be packaged and labeled as single bottles containing 30 OCA- or placebo-containing tablets, and should be dispensed to the subject

as instructed by the IWRS and according to the visit schedule in Table 1. Each bottle will be labeled with a unique bottle number. More than one bottle of investigational product may be dispensed to the subject at a visit to provide sufficient tablets for daily dosing until the next study visit.

For the LTSE period, investigational product will be packaged and labeled as single bottles containing 30 or 100 tablets of OCA and should be dispensed to the subject as instructed by the IWRS. Each bottle will be labeled with a unique bottle number. More than one bottle of investigational product may be dispensed to the subject at a visit to provide sufficient tablets for daily dosing until the next study visit.

## 10.3. Investigational Product Storage

Investigational product should be stored in the containers in which they are received from the Sponsor's supplier, at 15°C to 25°C.

## **10.4.** Investigational Product Administration

Subjects will begin dosing at the clinic following Randomization and will be instructed to take investigational product at approximately the same time each day with water. Subjects must be instructed to swallow one tablet whole; they must not chew, divide, or crush the tablet.

#### 10.4.1. Investigational Product Dispensation

On Randomization/Day 1, after confirmation of subject eligibility, the Investigator or designee will dispense investigational product to the subject. Before leaving the clinic, study site staff will ensure that the subject fully understands the dosing instructions.

Investigational product will be dispensed at clinic visits after confirmation of continued subject compliance and eligibility. If necessary, in exceptional circumstances, and only after approval by the Sponsor, investigational product may be delivered to subjects by courier, with proper precautions and documentation of shipping.

#### 10.4.2. Missed Doses

Subjects who miss a dose of investigational product should be instructed to take it later the same day, as soon as they remember. "Missed" doses should not be taken on a subsequent day (ie, the subject should not take more than the prescribed daily dose). Subjects will be asked to record the day they miss a dose.

#### 10.5. Atorvastatin Tablets

Atorvastatin tablets for oral administration contain 10 mg, 20 mg, and 40 mg atorvastatin and the following inactive ingredients: calcium carbonate, USP; candelilla wax, FCC; croscarmellose sodium, NF; hydroxypropyl cellulose, NF; lactose monohydrate, NF; magnesium stearate, NF; microcrystalline cellulose, NF; Opadry White YS-1-7040 (hypromellose, polyethylene glycol, talc, titanium dioxide); polysorbate 80, NF; simethicone emulsion.

#### 10.5.1. Atorvastatin Packaging and Labeling

Atorvastatin is commercially available and will be supplied as tablets in its commercial configuration, though all bottles will have an auxiliary label with study protocol number and bottle number for compliance. A designated vendor will be responsible for the distribution of atorvastatin to the Investigator.

Atorvastatin should be dispensed to the subject and dosed as instructed by the IWRS.

#### 10.5.1.1. Atorvastatin Storage

Atorvastatin should be stored in the containers in which they are received from the Sponsor's supplier, at the manufacturer's recommended storage conditions.

#### 10.5.2. Atorvastatin Administration

Subjects will be instructed to begin atorvastatin dosing on the day following their Week 4 Visit. The first dose will be administered at the study site during the subject's study visit (Table 1). Atorvastatin can be administered as a single dose with water at any time of the day, with or without food.

## 10.5.3. Atorvastatin Dispensation

At the subject's Week 4 Visit, the Investigator or designee will dispense a bottle containing atorvastatin 10-mg tablets to the subject. At the subject's Week 8 Visit, the Investigator or designee will dispense atorvastatin 10-mg tablets to the subject advising the subject to take 2 tablets for a total dose of atorvastatin 20 mg. At subsequent visits, atorvastatin will be dispensed as clinically indicated. For doses higher than 20 mg, subject may take multiple atorvastatin tablets for a total dose of 40 mg or 80 mg, as clinically indicated. Before leaving the clinic, study site staff will ensure that the subject fully understands the dosing instructions.

Upon confirmation of continued subject compliance and eligibility, atorvastatin will be dispensed using IWRS inventory management during study visits.

#### 10.5.4. Missed Doses of Atorvastatin

Subjects who miss a dose of atorvastatin should be instructed to take it later the same day, as soon as they remember. "Missed" doses should not be taken if it has been more than 12 hours since when they would normally take it; the next dose should be taken when they would normally dose. Subjects should be instructed not to take 2 doses at the same time. Subjects should be asked to record the day they miss a dose.

#### 10.5.5. Atorvastatin Overdose

There is no specific treatment for an overdose of atorvastatin. In the event of an overdose, the subject should be treated symptomatically, and supportive measures instituted as required. Due to extensive drug binding to plasma proteins, hemodialysis is not expected to significantly enhance atorvastatin clearance.

# 10.6. Investigational Product and Atorvastatin Accountability and Disposal

The Sponsor's representative will ship investigational product and atorvastatin to the study site under appropriate storage conditions. All shipments of investigational product and atorvastatin should be unpacked and the contents reviewed immediately upon receipt. If it is not possible to verify the contents immediately, they must be stored under the appropriate storage conditions until verification of the contents is possible (ideally, within 1 business day from receipt). The pharmacist or designee should verify the investigational product and atorvastatin against the shipment documentation. The pharmacist or designee should contact the Sponsor immediately to report any concerns regarding the shipment.

All investigational product and atorvastatin will be provided for use only in this study and is not to be used for any other purpose. The Investigator or designee will maintain a full record of investigational product and atorvastatin accountability, including records of individual subject dispensing and final return or disposition (as directed by the Sponsor).

The study monitor, also known as the Clinical Research Associate (CRA), will review accountability records against dispensed and in stock investigational product and atorvastatin during onsite monitoring visits, at study completion, and in the event of premature study termination. The CRA will retrieve documentation detailing and confirming the return or destruction of investigational product and atorvastatin.

#### 11. ASSESSMENT OF EFFICACY AND PHARMACOKINETICS

## 11.1. Efficacy Assessments

An overview of parameters supporting primary, secondary, and exploratory objectives of the study are summarized in Table 4. Samples for the assessment of efficacy variables will be collected according to the schedule of study procedures for the double-blind period (Table 1) and LTSE (Table 2). For a complete list of variables, please refer to Appendix A.

#### **Table 4: List of Planned Assessments**

The efficacy assessments supporting the primary, secondary, and exploratory objectives of the study are as follows:

| | Parameters |
|---|---|
| Primary Endpoints | |
| LDL metabolism | LDL cholesterol concentration, particle size, and particle concentration |
| Secondary Endpoints | |
| Lipoprotein metabolism | HDL cholesterol concentration, particle size and particle concentration; VLDL cholesterol concentration, particle size and particle concentration; TG and total cholesterol concentrations; ApoA1, ApoB, ApoE, ApoCII, ApoCIII and Lp(a) concentrations; PCSK9 concentration |
| Reverse cholesterol transport | Pre-β1 HDL concentration, macrophage cholesterol efflux; LCAT activity; CETP activity |
| <b>Exploratory Endpoints</b> | |
| Liver biochemistry and markers of liver function <sup>a</sup> | Albumin, ALP, ALT (isoenzymes), AST, direct bilirubin, GGT, INR, total bilirubin |
| Markers of liver inflammation | IL-6, hs-CRP, and TNF-α |
| Marker for hepatic apoptosis and fibrosis | CK-18-M30 and CK-18-M65 |
| Glycemic Control <sup>b</sup> | Glucose, insulin, C-peptide, HbA1c, HOMA-β, and HOMA-IR |
| OCA pharmacokinetics | OCA, tauro-OCA, glyco-OCA, total OCA, potentially other conjugates or metabolites not yet identified |
| Atorvastatin bioanalytical concentrations | Atorvastatin and its metabolites |
| Anthropometric measures <sup>c</sup> | Height, weight, and waist and hip circumference measurements; and BMI, and waist-to-hip ratio calculations |
| Pharmacodynamics | C4 (7α-hydroxy-4-cholesten-3-one) and FGF-19; possible analysis of conjugated and unconjugated bile acids |
| Noninvasive radiological liver fibrosis measurements | By TE (where available) |
| Cardiovascular risk scores | FRS and Reynolds scores |

ALP = alkaline phosphatase; ALT = alanine aminotransferase; ApoA1 = apolipoprotein A1; ApoB = apolipoprotein B; ApoCII = apolipoprotein CII; ApoCIII = apolipoprotein CIII; ApoE = apolipoprotein E; AST = aspartate aminotransferase; BMI = body mass index; C4 =  $7\alpha$ -hydroxy-4-cholesten-3-one; CK-18-M30 = cytokeratin-18 neoepitope M30; CK-18-M65 = cytokeratin-18 neoepitope M65; CTEP = cholesterol ester transfer protein; ECG = electrocardiogram; FGF-19 = fibroblast growth factor-19; FRS = Framingham Risk Score; GGT = gammaglutamyl transferase; HbA1c = hemoglobin-specific A1c fraction; HDL = high-density lipoprotein; HOMA- $\beta$  = homeostatic model assessment—beta-cell function, HOMA-IR = homeostatic model assessment – insulin resistance; hs-CRP = high-sensitivity C-reactive protein; IL-6 = interleukin-6; LCAT = lecithin cholesterol acyltransferase; LDL = low-density lipoprotein; Lp(a) = lipoprotein(a); PCSK9 = proprotein convertase subtilisin/kexin type 9;TE = transient elastography; TEAE = treatment-emergent adverse event; TG = triglycerides; TNF- $\alpha$  = tumor necrosis factor- $\alpha$ ; VLDL = very low-density lipoprotein

- <sup>a</sup> Liver biochemistry panel will be included in the serum biochemistry (see Table 10).
- <sup>b</sup> HOMA-IR is calculated from fasting plasma glucose and fasting serum insulin values.
- <sup>c</sup> Height will be measured at Screening only. BMI and waist-to-hip ratio will be calculated via EDC from waist and hip circumference measurements.

Please note that there are 2 distinct lipid assessments: the assessment of lipoprotein metabolism and the safety lipids assessment measured as part of serum chemistry. The latter will be used for randomization and safety assessments and the lipoprotein analysis samples will be used for the efficacy assessment.

#### 11.1.1. Efficacy Laboratory Assessments

The complete list of planned laboratory assessments supporting primary, secondary, and exploratory objectives of the study is shown in Table 4, and includes parameters related to LDL metabolism, lipoprotein metabolism, reverse cholesterol transport, liver biochemistry and markers of liver function, markers of inflammation, glycemic control, OCA PD markers, and NASH disease severity markers CK-18-M30 and CK-18-M65.

Fasting (8 hours) blood samples are required for efficacy analyses. During each visit, the Investigator or designee will verify that the subject has fasted for at least 8 hours and record fasting status in the source and eCRF. If the subject reports having eaten (water is permitted) within 8 hours, the Investigator or designee will document accordingly in the source and eCRF and remind the subject that fasting is required prior to onsite visits.

Blood samples will be collected at visits indicated in the Schedule of Study Procedures (Table 1 and Table 2).

#### 11.1.2. Liver Biopsy

Liver biopsy will be scheduled at Screening Visit 1 for confirmation of NASH (inclusion criteria) if no biopsy slides or tissue collected within 1 year of the Screening Visit 1 is available for central read. No other biopsy sample will be collected during the double-blind or LTSE phase of the study.

Biopsies should be at least 2 cm in length. All biopsies will be read centrally by a Sponsor-designated central reader.

#### 11.1.2.1. Central Reading of Liver Histology

Full instructions concerning the number and type of samples to be collected at each visit, the sample collection methods, sample processing, labeling, and shipping will be provided by the Sponsor in a study-specific histology manual.

All biopsy assessments, including determination of study eligibility based on NASH diagnosis and fibrosis staging during Screening, will be performed centrally by an independent pathologist. The central pathologist must confirm histological presence of NASH and a minimum NAS of 4 with a score of at least 1 in each component of NAS. Key features of NASH (ie, steatosis, lobular inflammation, and hepatocellular ballooning) will be graded in accordance with the NASH CRN criteria for scoring (Kleiner 2005) as summarized in Table 5. Fibrosis staging for eligibility will also be performed in accordance with NASH CRN criteria for fibrosis staging.

Table 5: NASH CRN Scoring System for Determining Eligibility and Primary Histological Endpoint Assessment

| NAFLD Activity Score (NAS) | | Fibrosis Staging | |
|---|---|---|---|
| Parameter | Scoring Criteria | Parameter | Staging Criteria |
| Steatosis | 0 = <5% $1 = 5% - 33%$ $2 = >33% - 66%$ $3 = >66%$ | Stage 0 | No Fibrosis |
| Lobular<br>Inflammation | 0 = No Foci<br>1 = <2 Foci per 200 × field<br>2 = 2 - 4 Foci per 200 × field<br>3 = >4 Foci per 200 × field | Stage 1<br>Stage 1a<br>Stage 1b<br>Stage 1c | Perisinusoidal or Periportal Mild, zone 3, perisinusoidal Moderate, zone 3, perisinusoidal Portal / periportal |
| Ballooning | 0 = None<br>1 = Few balloon cells<br>2 = Many cells / prominent ballooning | Stage 2 Stage 3 | Perisinusoidal and portal / periportal Bridging fibrosis |
| | 2 many const prominent ouncoming | Stage 4 | Cirrhosis |

In addition to the primary scoring system of NASH CRN, biopsy samples will also be scored based on modified Ishak scoring (Ishak 1995) for all subjects. Any extra biopsy tissue may undergo exploratory histological evaluations.

#### 11.1.3. Noninvasive Radiological Liver Fibrosis Measurements

Liver stiffness will be assessed during LTSE using a noninvasive radiological method TE at study sites where available.

#### 11.1.4. Blood Samples for Future Analysis

Blood samples for exploratory future analysis may be assessed for analytes such as adiponectin, plasminogen activator inhibitor-1(PAI-1), and B-type natriuretic peptide (BNP; Table 10). Blood samples may also be used to assess other disease or investigational product characteristics. The samples will be stored for up to 1 year after the end of the study and destroyed if not analyzed.

## 11.2. Pharmacokinetic and Pharmacodynamic Assessments

Parent OCA and its major conjugates (glyco-OCA and tauro-OCA), C4, and FGF-19 concentrations will be determined for OCA PK and FXR activity in OCA-treated subjects. Concentrations of atorvastatin and its metabolites will be assessed in PK sampled subjects. Samples will be obtained for possible assessment of conjugated and unconjugated bile acids.

#### 11.2.1. Pharmacodynamic Assessments

PD assessments will be collected according to the Schedule of Study Procedures (Table 1 and Table 2) from all subjects to measure C4, FGF-19, and possibly conjugated and unconjugated bile acids (dependent on the results of the C4 and FGF-19 assessments).

#### 11.2.2. Pharmacokinetic Assessments

Subjects who opt to participate in the PK assessment will provide blood samples for the measurement of OCA and its conjugates, and atorvastatin and its metabolites. The first sample should be collected within 30 minutes prior to administration of investigational product (predose) on Day 1 and prior to administration of investigational product or atorvastatin at the Week 16 Visit. Subjects will then receive a single dose of investigational product with approximately 240 mL of water. Serial blood samples will be obtained for measurement of OCA and its conjugates, and atorvastatin and its metabolites, at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until after the 1-hour sample is collected. A meal will be provided following collection of the 1-hour PK sample; the meal will be a meal replacement drink with nutrition information that has been submitted to and approved by the Sponsor in advance.

## 11.3. Anthropometric Assessments

Anthropometric measures include height (measured at Screening Visit 1 only), weight, and waist and hip circumference measurements. Waist-to-hip ratio will be calculated by the electronic data capture (EDC) system and will be calculated as ([Waist Circumference in Centimeters] / [Hip Circumference in Centimeters]). Height will also be collected at Screening Visit 1. Anthropometric measures will be performed during the visits indicated in Table 1 and Table 2.

#### 11.3.1. BMI

BMI will be calculated as (Weight in Kilograms / [Height in Meters × Height in Meters]). Instructions for measuring body weight and waist and hip circumference are described below. All three measures are to be obtained after the subject has fasted for at least 8 hours.

#### 11.3.2. Body Weight

Body weight should be obtained with the subject wearing a hospital gown or similar light clothing and no shoes, and with an empty bladder. The same scale should be used throughout the study. The floor surface on which the scale rests must be hard rather than carpeted or covered with other soft material. The subject should stand in the center of the platform. The weight is to be read and recorded to the first decimal point (eg. 97.1 kg) by study staff.

#### 11.3.3. Waist and Hip Circumference:

The subject should be wearing little clothing and standing upright during the measurements, with arms relaxed at the side, feet close together, and body weight evenly distributed. Waist circumference should be measured at the end of several consecutive natural breaths, midpoint between the top of the iliac crest and the lower margin of the last palpable rib in the mid-axillary line. Hip circumference should be measured at the largest circumference of the buttocks. Both measurements should be made with a Sponsor-provided measuring tape that is wrapped snugly around the subject, but not to the point that the tape is constricting. The tape must be level and parallel to the floor at the point of measurement. Each measurement should be repeated twice; if

the measurements are within 1 cm of one another, the average should be calculated. If the difference between the 2 measurements exceeds 1 cm, the 2 measurements should be repeated.

#### 12. ASSESSMENT OF SAFETY

Safety will be monitored and assessed by AEs/SAEs, medical history, physical examination, vital signs measurements, ECG results, and clinical laboratory assessments. Refer to Section 17.1 for AE reporting procedures.

#### 12.1. Adverse Events and Serious Adverse Events

#### 12.1.1. Definitions

#### **12.1.1.1.** Adverse Event

An AE is defined as any untoward medical occurrence associated with the use of the investigational product in humans, whether or not considered related to investigational product. An AE can be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with any use of the investigational product, without any judgment about causality and irrespective of route of administration, formulation, or dose, including an overdose. For this study, investigational product refers to OCA or placebo, and study medication refers to atorvastatin.

AEs include, but are not limited to: (1) a worsening or change in nature, severity, or frequency of condition(s) present at the start of the study; (2) subject deterioration due to primary illness; (3) intercurrent illness; and (4) drug interaction.

Subjects should be questioned in a general way, without leading the subject or asking about the occurrence of any specific symptom. The Investigator should attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. The diagnosis and not the individual signs/symptoms should be documented as the AE. For example, if the underlying disease process is a stroke, it would not be appropriate to record the AE by describing the symptoms "sudden numbness, dizziness, and difficulty speaking." The AE medical term of "stroke or cerebrovascular accident" should be recorded as it more accurately describes the AE.

#### 12.1.1.2. Treatment-Emergent Adverse Event

A treatment-emergent AE (TEAE) is any event not present before the initiation of the investigational product or any event already present that worsens in either intensity or frequency following exposure to the investigational product.

#### 12.1.1.3. Serious Adverse Event

An AE is considered 'serious' if, in the view of either the Investigator or Sponsor, it results in any of the following outcomes:

- Death
- Is immediately life threatening

• Requires in-patient hospitalization or prolongation of existing hospitalization

- Results in persistent or significant disability or incapacity
- Results in a congenital abnormality or birth defect
- Is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above

Events **not** considered to be SAEs are hospitalizations for:

- Routine monitoring of the studied indication and not associated with any deterioration in condition or AE;
- Elective treatment for a pre-existing condition that did not worsen;
- Respite care or observation when there is no AE associated with the hospitalization.

#### 12.1.2. Relationship to Investigational Product or Study Medication

The Investigator will document her/his opinion of the relationship of the AE to treatment with investigational product and study medication (atorvastatin) using the criteria outlined in Table 6. Each AE will be assessed for relationship to investigational product and atorvastatin independently. An AE for which there is a "reasonable possibility" that either investigational product or atorvastatin caused the AE is otherwise referred to as a suspected adverse reactions (SARs). "Reasonable possibility" means there is evidence to suggest a causal relationship between the investigational product and/or atorvastatin and the AE.

If the relationship between a SAE and the investigational product is determined to be "definite," "probable," or "possible," the event will be considered to be related to the investigational product for the purpose of assessing expedited regulatory reporting.

If the relationship between an SAE and the atorvastatin is determined to be "definite," "probable," or "possible," the event will be considered to be related to atorvastatin for the purpose of assessing expedited safety reporting and reporting to the manufacturer.

**Table 6:** Relationship of Adverse Events to Investigational Product or Study Medication

| Relationship | Description |
|---|---|
| Definite | A reaction that follows a reasonable temporal sequence from administration of the investigational product or study medication in which the investigational product or study medication level has been established in body fluids or tissue; that follows a known or expected response pattern to the suspected investigational product or study medication;; and that is confirmed by improvement on stopping or reducing the dosage of the investigational product or study medication, and reappearance of the reaction on repeated exposure. |
| Probable | A reaction that follows a reasonable temporal sequence from administration of the investigational product or study medication; that follows a known or expected response pattern to the suspected investigational product or study medication; that is confirmed by stopping or reducing the dosage of the investigational product or study medication; and that could not be reasonably explained by the known characteristics of the subject's clinical state. |
| Possible | A reaction that follows a reasonable temporal sequence from administration of the investigational product or study medication; that follows a known or expected response pattern to the suspected investigational product or study medication; but that could readily be produced by a number of other factors. |
| Unlikely | An event that does not follow a reasonable temporal sequence from administration of the investigational product or study medication; that does not follow a known or suspected response pattern to the suspected investigational product or study medication; and that could reasonably be explained by known characteristics of the subject's clinical state. |
| Not Related | Any event that does not meet the above criteria. |

#### 12.1.3. Relationship to Liver Biopsy

The Investigator will document her/his opinion of the relationship of the AE to liver biopsy using the criteria outlined in Table 7.

**Table 7:** Relationship of Adverse Events to Liver Biopsy

| Relationship | Description |
|---|---|
| Definite | A reaction that follows a reasonable temporal sequence from the liver biopsy, and that follows a known or expected response pattern to the liver biopsy. |
| Not Related | Any event that does not meet the above criteria. |

#### 12.1.4. Recording Adverse Event Severity

AEs must be graded for severity (ie, intensity) using Common Terminology Criteria for Adverse Events (CTCE) Version 4.03 (Appendix C). A severity category of mild, moderate, severe, life-threatening, or death as defined in Table 8, must be entered on the AE eCRF. It should be noted that the term "severe" used to grade intensity is not synonymous with the term "serious." The assessment of severity is made regardless of investigational product relationship or of the seriousness of the AE. When reporting AEs, reference should be made to the CTCAE manual for guidance on appropriate grading.

**Table 8:** Severity of Adverse Events

| Grade | Clinical Description of Severity |
|---|---|
| 1 = Mild | Asymptomatic or mild symptoms, clinical or diagnostic observations only, or intervention not indicated. |
| 2 = Moderate | Minimal, local or noninvasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. <sup>a</sup> |
| 3 = Severe | Medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, or limiting self-care activities of daily living. <sup>b</sup> |
| 4 = Life-<br>Threatening | Urgent intervention indicated |
| 5 = Death | Death related to AE |

<sup>&</sup>lt;sup>a</sup> Instrumental activities of daily living refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

## 12.1.4.1. Severity of Pruritus (as an AE)

Pruritus was the most common AE seen in the Phase 2 PBC studies of OCA and thus may occur in this study.

To ensure consistency in reporting, the following guidelines for assessing severity of pruritus should be used for AE reporting. As pruritus is a subjective symptom, clinical judgment should be used to determine its severity and management (Table 9).

**Table 9:** Severity of Pruritus

| Pruritus Grade | Clinical Description of Severity for Pruritus and Medical Intervention |
|---|---|
| 1 = Mild | Generally localized; causing no limitation of usual activities or minimal sleep disturbance; the subject may experience slight discomfort. Medicinal intervention is not indicated. |
| 2 = Moderate | Intense or widespread; causing some limitation of usual activities or sleep disturbance; the subject may experience annoying discomfort. Medicinal intervention may be indicated. |
| 3 = Severe | Intense or widespread and interfering with activities of daily living, ie, causing inability to carry out usual activities, or severe sleep disturbance; the subject may experience intolerable discomfort. Medicinal intervention is typically indicated. |

Since pruritus is a subjective symptom and the occurrence and magnitude of which are not readily measured by objective tools, clinical judgment needs to be applied in the management of each subject. Managing OCA-related pruritus may help improve tolerance in those subjects who experience problematic pruritus and may otherwise discontinue from the study prematurely. General guidance for the management of subjects experiencing significant pruritus includes:

<sup>&</sup>lt;sup>b</sup> Self-care activities of daily living refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

• Drug holiday: A drug holiday is defined as an Investigator 'prescribed' complete interruption of dosing for 1 or more consecutive days (ie, non-daily dosing does not constitute a drug holiday). Details of drug holidays and/or nondaily dosing regimens should be recorded in the CRF. Per Section 8.4.1.1, subjects with pruritus ≥Grade 3 in severity and possibly, probably, or definitely related to investigational product must discontinue investigational product.

- Prescribe BAS. Subjects taking BAS (including colestyramine and its derivatives, colestipol, colesevelam, or other sequestrants) should be instructed to stagger their dosing of investigational product, ensuring at least 4 hours between doses of the BAS and investigational product.
- Other therapies may be tried as deemed clinically appropriate.
- Less frequent dosing of investigational product (eg, on alternate days) may be tried, after which subjects may return to their original daily dose as soon as tolerated.

#### 12.1.5. Reporting of Adverse Events and Serious Adverse Events

#### 12.1.5.1. Reporting of Adverse Events

AE data will be collected from the time that signed informed consent is obtained until the subject fully completes her/his study participation.

All AEs, whether believed by the Investigator to be related or unrelated to the investigational product, must be documented in the subject's medical records, in accordance with the Investigator's normal clinical practice and in the eCRF in the EDC system. Each AE is to be evaluated for duration, intensity, frequency, seriousness, outcome, other actions taken, and relationship to the investigational product or study medication.

#### 12.1.5.2. Reporting of Serious Adverse Events

In agreeing to the provisions of this protocol, the Investigator accepts all legal responsibilities for immediate reporting of SAEs to the Sponsor. Immediate reporting implies within 24 hours of becoming aware of the occurrence of an SAE.

All SAEs must be reported to the Sponsor. SAEs are reported by entering the SAE data into the study specific EDC system. Entering the SAE data into the EDC system will automatically notify the Sponsor of the event. In the event that the EDC system is inaccessible, an SAE may be reported by:

- E-mail to the SAE email address: sae@interceptpharma.com
- Fax using a paper SAE report form: +1 800 497 8521
- Telephone: +1 844 250 6396

If an SAE is reported by telephone or fax, an SAE Report form must also be completed in the EDC system as soon as the EDC system is accessible. At a minimum, the following information should be provided at the time of the initial report:

- Subject number
- Event term
- At least 1 criterion classifying the event as serious
- Name and title of the reporting individual
- Causal relationship to the investigational product or study medication

The Investigator will assess whether the event is causally related to the investigational product or study medication. The Sponsor will also assess whether the event is causally related to the investigational product, in addition to assessing the overall safety profile of the investigational product. The Sponsor will notify the appropriate regulatory agencies as well as all participating Investigators of investigational new drug (IND) Safety Reports/Expedited Safety Reports that occur during the study within the time frames required by each regulatory agency.

Following the initial report, any additional information obtained by the Investigator about the SAE must be reported promptly to the Sponsor in the same manner as described above for the initial SAE report. Any supporting source documentation should be faxed to +1 800 497 8521 or emailed to sae@interceptpharma.com as soon as possible.

The Investigator is responsible for submitting information on IND Safety Reports/Expedited Safety Reports received from the Sponsor to her/his local IRB/IEC, as directed by the local country requirements.

Documentation of the submissions to IRBs/IECs must be retained in the appropriate study file(s). As instructed by the Sponsor, IND Safety Reports/Expedited Safety Reports should be retained in the appropriate investigative site study files, or with the IB.

#### 12.1.6. Additional Investigator Responsibilities for SAEs

The safety data recorded in the EDC represent the official record of all AEs and SAEs reported in the study. The Investigator should comply with requests by the Medical Monitor or other Sponsor personnel to record the SAE on the subject's AE eCRF in the EDC. Other supporting documents such as radiology reports, hospital discharge summaries, and autopsy reports should also be provided, when appropriate. Additionally, upon request by the Sponsor, the Investigator should provide input into the SAE narrative and provide timely information to ensure prompt follow-up and closure of the SAE report.

The Investigator and supporting personnel responsible for subject care should discuss with the Medical Monitor any need for supplemental investigations of SAEs. The results of these additional assessments must be reported to the Medical Monitor.

#### 12.1.7. Notification of Post-Study SAEs

If an Investigator becomes aware of an SAE that may be attributable to the investigational product at any time after the end of the study, the Sponsor should be notified immediately (ie, within 24 hours).

All SAEs that occur within 30 days following the cessation of investigational product or study medication, whether or not they are related to the study, must be reported to the Sponsor within 24 hours by following the instructions provided in Section 12.1.5.2.

#### 12.1.8. Follow-Up of Adverse Events and Serious Adverse Events

All AEs must be followed during the course of the study until the AE resolves, is no longer of clinical concern, has stabilized or is otherwise explained, or the subject is lost to follow-up.

AEs ongoing at the final visit that are deemed to be "possibly, probably, or definitely" related or of other clinical significance must be followed for as long as necessary to adequately evaluate the safety of the subject or until the event stabilizes, resolves, or is no longer of clinical concern. If resolved, a resolution date for the AE should be documented in the EDC. The Investigator must ensure that follow-up includes any supplemental investigations indicated to elucidate the nature and/or causality of the AE. This may include additional laboratory tests or investigations, or consultation with other healthcare professionals, as considered clinically appropriate by the Investigator.

All subjects showing possible drug-induced liver injury should be followed until all abnormalities return to normal or to the baseline state. Drug-induced liver injury may develop or progress even after the causative drug has been stopped. Results should be recorded in the CRF. Note that longer follow-up can sometimes reveal an off-drug repetition of what had appeared to be drug-induced liver injury, indicating that liver injury was related to underlying liver disease.

#### 12.1.8.1. Pregnancy and Follow-Up

Pregnancies are not considered AEs in and of themselves; however, if a female study participant becomes pregnant while she is enrolled in the clinical study, she must discontinue treatment with investigational product and atorvastatin immediately (see Section 8.4.1.1) and the Sponsor must be notified within 24 hours of the Investigator's awareness of the pregnancy by completing the Pregnancy eCRF in the EDC system and downloading and completing the Pregnancy Report Form. The Pregnancy Report Form must be emailed to sae@interceptpharma.com or faxed to +1-800-497-8521. The subject and neonate must be followed for outcome information and/or as considered appropriate by the Investigator and the Sponsor.

Women who discontinue the study due to pregnancy may not re-enroll in the study at any point, but should continue with the study visit schedule and must be followed by the Investigator through pregnancy outcome. Similarly, if a subject's pregnancy is terminated early (planned or unplanned), the subject will also be removed from the study.

Completing the Pregnancy Report Form is not a substitute for reporting an AE/SAE if an AE/SAE has occurred related to or concurrent with the pregnancy. In the situation when an AE/SAE has occurred, the AE/SAE reporting procedures described in Section 17.1 must also be followed.

## 12.2. Other Safety Parameters

#### 12.2.1. Medical History/Demographics

A complete medical history will be obtained from the subject at Screening Visit 1. Alcohol consumption history will be recorded. Demographic characteristics (age, gender, race, and ethnicity) will be recorded.

#### 12.2.2. Physical Examination

To assess for clinical findings, the Investigator or designee will perform a physical examination at the timepoints specified in the Schedule of Study Procedures (Table 1 and Table 2). This includes height, which is only measured and recorded at Screening Visit 1. The physical examination must include the following:

- General appearance
- Height (Screening Visit 1 only)
- Weight (and BMI, if applicable)
- Skin
- Head, eyes, ears, nose, and throat
- Neck
- Lymph nodes
- Chest/Respiratory system
- Cardiovascular system
- Abdominal region
- Extremities
- Musculoskeletal system
- Mental status
- Neurological system

#### 12.2.3. Vital Signs

Vital signs will be assessed at indicated visits (Table 1 and Table 2). Vital signs include body temperature, sitting heart rate, respiratory rate, and sitting blood pressure. When taking heart rate, respiratory rate, and blood pressure readings, subjects should be seated quietly for a minimum of 3 minutes before the readings are taken.

#### 12.2.4. Electrocardiogram

Standard 12-lead ECGs will be collected at the visits specified in Table 1 and Table 2. The Investigator or designee will review the 12-lead ECG and findings will be recorded in the eCRF as normal, abnormal but not clinically significant, or abnormal and clinically significant. Any

clinically significant abnormalities on ECGs recorded after Randomization/Day 1 will also be documented as AEs and entered on the AE page of the eCRF, whereas abnormalities on ECGs up to Randomization/Day 1, prior to administration of the investigational product, will be recorded as pre-treatment AEs.

Investigative sites must retain a copy of all 12-lead ECGs evaluated by the Investigator or designee. These ECGs must be clearly labeled with the Subject ID number, date, and time. Full instructions will be provided for forwarding the 12-lead ECGs for central reading.

#### 12.2.5. Alcohol Consumption

Information about the subject's alcohol consumption will be collected during the visits indicated in Table 1 and Table 2 using the Alcohol Use Disorders Identification Test (AUDIT). AUDIT is a 10-item questionnaire that uses the domains of alcohol consumption, drinking behavior, and alcohol-related problems (Saunders 1993).

#### 12.2.6. Laboratory Assessments

Except for Screening Visit 1, subjects will be instructed to attend each study visit in a fasted state, and subjects should remain fasted until their blood samples have been collected. For visits that require fasting, the Investigator or designee will verify that the subject has fasted for at least 8 hours and record fasting status in the source and eCRF. If the subject reports having eaten (water is permitted) within the past 8 hours, the Investigator or designee will document accordingly in the source and eCRF and remind the subject that fasting is required before all study visits (see Section 9.6.1).

Blood, and urine samples for laboratory assessments will be collected at the visits specified in Table 1 and Table 2. Full instructions concerning the number and type of samples to be collected at each visit, the required sample volumes, sample collection methods, sample processing, labeling, and shipping will be provided in a separate procedural manual. All necessary collection supplies will be provided by the central laboratory and will be appropriately assembled for the specific evaluations required at each visit.

The list of laboratory analytes to be tested is shown in Table 10.

**Table 10:** List of Laboratory Analytes to be Tested

| Laboratory Assessment | Analyte |
|---|---|
| All Subjects | |
| Serum chemistry | Albumin, BUN, creatinine, conjugated (direct) bilirubin, total bilirubin, AST, ALT, ALP (isoenzymes), GGT, creatine phosphokinase, electrolytes (calcium, chloride, magnesium, phosphorus, potassium, sodium), total protein, bicarbonate, free fatty acids; and blood lipids (total cholesterol, LDL, HDL, and VLDL fractions and TGs) |
| Hematology | Hemoglobin, hematocrit, white blood count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelets, red blood cell count (including MCV, MCH, MCHC) |
| Urinalysis | pH, specific gravity, protein, glucose, ketones, bilirubin, blood, microscopic exam |
| Coagulation | PT, PTT, INR |
| Glycemic control measures | Fasting plasma glucose, insulin, C-peptide, HbA1c, HOMA-β, and HOMA-IR |
| Lipoprotein analysis <sup>a</sup> | LDL, HDL, VLDL, total cholesterol, triglycerides, ApoA1, ApoB, ApoE, ApoCII, ApoCIII and Lp(a), PCSK9 |
| Reverse Cholesterol Transport | Pre-β HDL, macrophage cholesterol efflux, LCAT and CETP |
| Markers of Inflammation | IL-6, hs-CRP, and TNF-α |
| Markers of fibrosis and apoptosis | CK-18-M30 and CK-18-M65 |
| Vitamin D levels | Vitamin D |
| Thyroid function tests | T3, T4, TSH |
| PD Assessment | C4 and FGF-19; possible analysis of conjugated and unconjugated bile acids |
| Blood sample for future analysis, including markers of cardiovascular risk | Adiponectin, PAI-1, BNP |
| Pregnancy Test (female subjects of childbearing potential) | β-hCG |
| Virus screening tests | Hepatitis B surface antigen, hepatitis C antibody, and HCV ribonucleic acid [RNA] |
| Subset of Subjects | |
| PK analytes | OCA, tauro-OCA, glyco-OCA, and possible other conjugates or metabolites not yet identified Atorvastatin and its metabolites |

ALP = alkaline phosphatase; ALT = alanine aminotransferase; ApoA1 = apolipoprotein A1; ApoB = apolipoprotein B; ApoCI = apolipoprotein CI; ApoCII = apolipoprotein CII; ApoE = apolipoprotein E; AST = aspartate aminotransferase; BNP = B-type natriuretic peptide; BUN = blood urea nitrogen; C4 = 7α-hydroxy-4-cholesten-3-one; CETP = cholesterol ester transfer protein; CK -18-M30 = cytokeratin-18 neoepitope M30; CK-18-M65 = cytokeratin-18 neoepitope M65; GGT = gamma-glutamyl transferase; HbA1c = hemoglobin-specific

A1c fraction; HDL = high-density lipoprotein; HOMA- $\beta$  = homeostatic model assessment-beta-cell function; HOMA-IR = homeostatic model assessment – insulin resistance; hs-CRP = high-sensitivity C-reactive protein; IL-6 = interleukin-6; INR = international normalized ratio; LCAT = lecithin cholesterol acyltransferase; LDL = low-density lipoprotein; Lp(a) = lipoprotein(a); MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = mean corpuscular volume; PAI-1 = plasminogen activator inhibitor-1; PCSK9 = proprotein convertase subtilisin/kexin type 9; PK = pharmacokinetic; PT = prothrombin time; PTT = partial thromboplastin time; Pre- $\beta$ -HDL = pre- $\beta$ -high-density lipoprotein; TGs = triglycerides; T3 = triiodothyronine; T4 = thyroxine; TNF- $\alpha$  = tumor necrosis factor- $\alpha$ ; TSH = thyroid-stimulating hormone; VLDL = very low-density lipoprotein

<sup>a</sup> NMR-based panel will be used for LDL, HDL, and VLDL cholesterol concentrations, particle sizes, and particle concentrations. ApoA1, ApoB, ApoE, ApoCII, ApoCIII Lp(a), and PCSK9 concentrations will be measured using appropriate methods at central or specialty laboratories. Serum chemistry panel will be used for LDL, HDL, VLDL, TG, and total cholesterol concentration.

All subjects with laboratory tests containing clinically significant abnormal values are to be followed regularly until the values return to normal ranges; until a valid reason, other than investigational product related AE, is identified; or until further follow-up is deemed medically unnecessary.

The Investigator should manage subjects with clinically significant lipoprotein abnormalities using local standard of care procedures as appropriate after assessing the individual subject's total cardiovascular risk profile.

Urine-based  $\beta$ -hCG pregnancy tests will be performed for female subjects of childbearing potential at the visits specified in Table 1 and Table 2. If a urine pregnancy test is positive, a serum pregnancy test must be performed to confirm the result (Table 1, Table 2, and Section 9.7). If positive, the Sponsor must be notified and the subject will be followed, as outlined in Section 12.1.8.1 through pregnancy outcome.

International normalized ratio (INR) will be calculated based on prothrombin time value by the central laboratory. HOMA-IR values will be calculated based on fasting plasma glucose and insulin concentrations. Total OCA will be calculated based on OCA, tauro-OCA, and glyco-OCA concentrations.

#### 13. STATISTICS

## 13.1. Analysis Sets

The following subject populations will be used for presentation and analysis of data:

- <u>Intent-to-Treat (ITT) Population</u>: All randomized subjects who receive any amount of investigational product will be included in the ITT Population. Treatment assignment will be based on the randomized treatment allocation.
- <u>Safety Population</u>: The Safety Population will include all subjects who receive any amount of investigational product. Treatment assignment will be based on the treatment actually received. The Safety Population will be used for the analysis of all safety data.
- <u>Efficacy Evaluable Population</u>: All subjects who complete the double-blind phase according to the indicated doses of investigational product and atorvastatin without

any significant protocol deviations. The Efficacy Evaluable Population will be the primary population used for efficacy analyses.

- Pharmacokinetic Populations: The OCA PK Population will include all OCA subjects who consent to participate in the PK assessments and have at least one confirmed fasted analyzable sample. Subjects must have been fasting for approximately 8 hours before the visit and must not have any major protocol deviations that potentially affect exposure levels. The Atorvastatin PK Population will include all subjects who consent to participate in the PK assessments and have at least one confirmed fasted analyzable sample.
- <u>LTSE Population</u>: All subjects who receive any amount of investigational product as part of the LTSE will be included in the LTSE Population.

## **13.2.** Determination of Sample Size

It is the intent of this study to characterize the components of LDL metabolism (cholesterol concentration, particle size, particle concentration) in subjects with NASH before and after treatment with OCA and to assess the changes induced by HMG Coenzyme A reductase inhibitor (atorvastatin) therapy. Assuming, 22 mg/dL increase from baseline with a standard deviation of 24 in LDLc in the OCA 25 mg group without atorvastatin therapy after 16 weeks of treatment based on data from FLINT, a sample size of 20 subjects per group will provide greater than 97.3% power to demonstrate the statistically significant difference of LDLc increase from baseline with a 2-sided type I error of 0.05.

#### 13.3. General Statistical Considerations

A Statistical Analysis Plan (SAP), providing details about the specific planned analyses and statistical tests for both the double-blind phase and the LTSE phase, will be prepared and approved by the Sponsor and its designees prior to study database lock.

## 13.4. Handling of Dropout and Missing Data

Primary analysis of efficacy endpoints will be done using observed data only; missing values will not be imputed. A sensitivity analysis using a last observation carried forward approach may be considered.

## 13.5. Subject Population and Demographic Characteristics

Approximately 80 subjects with a confirmed diagnosis of NASH will be randomized to receive investigational product. Demographic characteristics including age, gender, race, and ethnicity will be summarized descriptively.

## 13.6. Efficacy Analysis

All efficacy analyses will be conducted using the Efficacy Evaluable Population. In addition, the ITT Population will be used for sensitivity analysis of the primary analyses.

The baseline value for efficacy analyses is defined as the last value prior to administration of investigational product on Day 1 (predose).

## 13.6.1. Primary Efficacy Analysis

The primary efficacy analysis, changes in LDL cholesterol, particle size and particle concentration at Week 16 (end of double-blind phase) compared to Baseline will be summarized by treatment group.

Analyses of observed values will be carried out using an analysis of covariance (ANCOVA) model at each visit with change from baseline as the dependent variable, including treatment group and randomization stratification factor as fixed effects and baseline as a covariate. The same analysis will be carried out using percentage change from baseline as the dependent variable.

Descriptive statistics of the values will be summarized by treatment group and visit. The results, change from baseline, and percentage change from baseline values as well as estimates of least-square (LS) means, standard errors, and 95% confidence intervals (CIs) will be presented by treatment group.

The comparison of LDLc change from baseline and percentage change from baseline values between each active treatment group and placebo group will be performed as exploratory analysis. Estimates of the LS mean difference between each active treatment group and placebo group, the standard error of the difference, and 95% CI of the difference will be presented.

Sensitivity analysis for primary efficacy analysis will be performed using the ITT Population.

#### 13.6.2. Secondary Efficacy Analysis

The secondary efficacy parameters will be analyzed in the same manner as the primary efficacy variables. Descriptive statistics will be generated and will include change from baseline, percentage change from baseline, and estimates of LS means, standard errors, and 95% CIs presented by treatment group.

The secondary parameters related to lipoprotein metabolism include HDL cholesterol concentration, particle size and particle concentration; VLDL cholesterol concentration, particle size and particle concentration; TG and total cholesterol concentrations; and ApoA1, ApoB, ApoEI, ApoCII, ApoCIII and Lp(a) concentrations.

The secondary parameters related to reverse cholesterol metabolism include pre-β1 HDL concentration, macrophage cholesterol efflux, lecithin cholesterol acyltransferase (LCAT) activity, cholesterol ester transfer protein (CETP) activity, and proprotein convertase subtilisin/kexin type 9 (PCSK9) enzyme levels.

#### 13.6.3. Additional Exploratory Efficacy Analyses

#### 13.6.3.1. Liver Biochemistry, Hepatobiliary Damage, and Liver Function

The following laboratory parameters will be summarized by treatment group: ALT, AST, gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), total and conjugated (direct) bilirubin, albumin, INR, and platelets.

Analyses of observed laboratory values will be carried out using an ANCOVA model at each visit with change from baseline as the dependent variable, including treatment group and randomization stratification factor as fixed effects and baseline as a covariate. The same analysis will be carried out using percentage change from baseline as the dependent variable.

Descriptive statistics will be used to summarize the laboratory values by treatment group and visit. The results, change from baseline, and percentage change from baseline; as well as estimates of LS means, standard errors, and 95% CIs will be presented by treatment group. Estimates of the mean difference between each active treatment group and placebo group, the standard error of the difference, and 95% CI of the difference will be presented.

#### 13.6.3.2. Markers of Inflammation, Fibrosis, and/or Apoptosis

Markers of hepatic fibrosis, inflammation, and/or apoptosis include IL-6, hs-CRP, TNF-α, and CK-18-M30 and CK-18-M65. These biomarkers will be summarized by treatment group using descriptive statistics at Baseline and at each post-Baseline visit. The absolute and percentage change from baseline will be analyzed using the Wilcoxon Rank Sum Test to compare treatment groups. The median differences and 95% CI of the median differences between treatment groups will be constructed using a Hodges-Lehmann estimate. If the median differences between treatments are not symmetrical around the median, the Sign Test may be used.

#### 13.6.3.3. Glycemic Control Measures

Glycemic control measures include fasting glucose, fasting insulin, C-peptide, HbA1c, HOMA-β, and HOMA-IR. These measures will be summarized by treatment group using descriptive statistics at Baseline and at each on-study evaluation. The change from baseline will also be summarized. Baseline is defined as the last fasting assessment prior to treatment. Treatment groups will be compared using an ANCOVA model at each visit with change from baseline as the dependent variable, including treatment group and randomization stratification factor as fixed effects and baseline as a covariate. The same analysis will be carried out using percentage change from baseline as the dependent variable. Estimates of LS means, standard errors, and 95% CIs will be presented by treatment group. Estimates of the mean difference between each active treatment group and placebo group, the standard error of the difference, and 95% CI of the difference will be presented. The distribution of glycemic control measures will be evaluated for normality assumptions. If normality assumptions are violated, non-parametric methods, such as a rank ANCOVA model, will be used.

Subgroup analyses will also be presented by diabetes status, excluding the randomization stratification factor from the ANCOVA model.

#### 13.6.3.4. Anthropometric Measures and Blood Pressure

Anthropometric measures include height (measured and recorded only at Screening Visit 1), body weight, and waist and hip circumference measurements; and BMI and waist-to-hip ratio calculations. Anthropometric and blood pressure measures will be summarized by treatment group using descriptive statistics at Baseline and at each on-study evaluation. The change from Baseline will also be summarized. Baseline is defined as the last assessment prior to treatment. Treatment groups will be compared using an ANCOVA model at each visit with change from

baseline as the dependent variable, including treatment group and randomization stratification factor as fixed effects and baseline as a covariate. The same analysis will be carried out using percentage change from baseline as the dependent variable. Estimates of LS means, standard errors, and 95% CIs will be presented by treatment group. Estimates of the mean difference between each active treatment group and placebo group, the standard error of the difference, and 95% CI of the difference will be presented.

Subgroup analyses will also be presented by diabetes status, excluding the randomization stratification factor from the ANCOVA model. Subgroup analyses of blood pressure will also be presented by use of antihypertensive medications.

#### 13.6.3.5. Noninvasive Radiological Liver Fibrosis Measurements

Noninvasive radiological methods to assess liver stiffness will be conducted at selected centers where the devices are available. These assessments include TE. Measurements (based on available data) will be summarized by treatment group using descriptive statistics at Baseline and at each post-Baseline Visit. The proportion of fibrosis improvement based on TE measurement will be summarized by treatment group at Week 16 of the double-blind phase, and year 1 and year 2 of the LTSE phase. The correlation with histological assessment based on biopsy at Baseline will also be assessed.

#### 13.6.3.6. Pharmacodynamic Analysis

C4, FGF-19, conjugated and unconjugated bile acids, and total bile acids will be summarized by treatment group using descriptive statistics at Baseline and at each scheduled post-Baseline Visit. The absolute change from baseline will also be summarized. Baseline is defined as the mean of all available evaluations prior to treatment.

#### 13.6.3.7. Pharmacokinetic Analysis

The PK Population will be used for analysis of PK parameters, which include plasma OCA (parent) and its conjugates (glyco-OCA and tauro-OCA), total OCA, atorvastatin and its metabolites, and potentially other analytes not yet identified. PK analysis will be conducted using standard non-compartmental methodologies.

For the analysis of OCA and its conjugates, values will be summarized by active treatment group using descriptive statistics. Only samples that have a confirmed fasting of approximately 8 hours or more before their visit will be included in the analysis.

Further details regarding the methods for calculating PK and the specific parameters to be reported will be described in the SAP.

#### 13.6.3.8. Cardiovascular Risk Scores

The cardiovascular risk score includes the FRS and Reynolds scores. Each score is derived from a subject's age, sex, smoking status, total cholesterol and HDL levels, and other factors including family history, BMI, ethnicity, and medications. Cardiovascular scores will be calculated at the time of data analysis. These markers will be summarized by treatment group using descriptive

statistics at Baseline and at each on-study evaluation. The change and percentage change from Baseline will also be summarized.

#### 13.6.4. LTSE Analyses

Similar analyses to that which are described above will be conducted for the LTSE using the double-blind baseline value. Analyses based on the double-blind baseline will be performed using randomized treatment groups (placebo, OCA 5 mg, OCA 10 mg, or OCA 25 mg). Sensitivity analyses may be conducted using the last value prior to first dose in the LTSE for all subjects.

## 13.7. Safety Analysis

Safety data, including AEs and clinical laboratory observations, will be summarized by treatment group using the Safety Population. The evaluation of safety data will be conducted for both the end of double-blind phase and final analyses at the end of the LTSE.

#### 13.7.1. Adverse Events

AEs will be coded using the Medical Dictionary of Regulatory Activities (MedDRA). Summary tables of TEAEs will be provided. The incidence of TEAEs and SAEs will be tabulated by system organ class and preferred term for each treatment group, and by severity and relationship to treatment. Tables of TEAEs leading to investigational product discontinuation and SAEs will be provided. The incidence of pre-treatment AEs and pre-treatment SAEs occurring after ICF signoff and before the first dosing of investigational product (OCA or placebo) will be tabulated in the same manner as above for all subjects participating in the washout period.

#### 13.7.2. Clinical Laboratory Evaluations

Laboratory parameters will be summarized by treatment group using descriptive statistics at Baseline and at each scheduled post-Baseline Visit. The absolute change from Baseline will also be summarized. Baseline is defined as the mean of all available evaluations (using fasting blood sample values for lipids and glucose) prior to treatment.

In addition, shift tables (ie, low-normal-high at Baseline versus low-normal-high at post-Baseline Visit in a 3-by-3 contingency table) from Baseline to worst value, last value, and at each scheduled post-Baseline Visit will be provided for hematology, coagulation, and serum chemistry by treatment group to assess changes in laboratory values from Baseline to each on-study evaluation.

#### 13.7.3. Lipoprotein Evaluations

Serum chemistry based assessments are the standard safety tool for monitoring subjects' serum lipids. Baseline is defined as the last fasting assessment prior to treatment. This analysis will only include samples that have a confirmed fasting of approximately 8 hours or more prior to the visit at which they were collected. Further analyses of lipoprotein analytes will be specified in the SAP.

Subgroup analyses will also be presented by use of statin medication.

#### 13.7.4. Additional Safety Analysis

#### **13.7.4.1.** Vital Signs

The results and change from baseline to each on-study evaluation visit will be summarized for body temperature, sitting heart rate, and respiratory rate.

#### 13.7.4.2. Electrocardiograms

The ECG data analysis will be conducted based on methodology recommended in the International Conference on Harmonisation (ICH) E14 guideline, The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Nonantiarrhythmic Drugs.

Baseline is defined as the mean of all available evaluations prior to treatment. Descriptive statistics of ECG parameters (time between 2 consecutive R waves [RR], PR, QRS, QT, and QT interval corrected by Fridericia's formula [QTcF]) at baseline and at each post-baseline timepoint will be summarized by treatment group; absolute changes from baseline will also be summarized.

A categorical summary of abnormal QTcF values will be presented by treatment group. The number of patients with values of >450 msec, >480 msec, and >500 msec will be presented, and the number of patients with change from baseline values of >30 msec and >60 msec will also be presented.

Overall interpretation results for ECGs and the Investigator interpretation results are collected as normal, abnormal not clinically significant, and abnormal clinically significant. Subjects whose interpretation shifts from normal to abnormal will be listed separately including description of the abnormality and any associated comments.

#### 13.7.5. Adjudicated Cardiovascular Events

Adjudicated cardiovascular events include core major adverse cardiovascular events (MACE; cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke) and expanded MACE (unstable angina requiring hospitalization, transient ischemic attack, peripheral or coronary revascularization procedures, hospitalization for congestive heart failure). Other events potentially related to adverse cardiovascular outcomes are defined in Appendix D and will be included in the Cardiovascular Adjudication Committee (CAC) Charter for adjudication. Undetermined cause of death will be classified as a cardiovascular death by the CAC.

Summaries of adjudicated cardiovascular events will include the incidence of TEAEs and the incidence of serious TEAEs. All summaries of incidence will include the associated exact binomial 95% CI.

## 13.8. Data Monitoring Committee

An independent DMC that includes hepatologists, pharmaceutical physicians, epidemiology/cardiology expert(s), and statistician(s) not involved in the study as Investigators, or consultants. The DMC will have oversight over the study conduct as defined by the DMC charter. All members will have considerable experience with clinical study conduct and DMCs. Any candidate found to have a conflict of interest or whose name is listed on the FDA debarment

list will not be offered membership. Conflicts of interest will be assessed regularly, and if members are found to have a new conflict of interest they would be replaced.

The DMC will meet approximately quarterly at scheduled meetings and ad hoc meetings will be convened, as appropriate, to review safety and efficacy data. Based on review of these data, the DMC will advise the Sponsor on the validity and scientific merit of continuing the study.

Written minutes of both the open and closed DMC sessions will be prepared. The closed minutes will be made available to the appointed Sponsor representatives only after the double-blind database is locked and unblinded.

Data listings provided to the DMC do not contain individual subject treatment information; however, the DMC will have access to the database and may unblind individual subject data as appropriate. Summary tables reviewed by the DMC during closed sessions will include an overall column containing information regarding all subjects and separate treatment columns with fake labels, ie, the actual treatment groups are used, but are not identified. Data reviewed during the meetings will include, at a minimum, disposition, demographics, exposure, clinical laboratory results, MedDRA coded AEs, and AEs leading to early withdrawal of investigational product. At each meeting, detailed narratives of interval SAEs (including events resulting in death) are reviewed by the DMC in addition to a cumulative list of all SAEs.

The DMC may agree to adjust meeting frequency based upon actual and projected safety and efficacy data availability.

All Investigators and responsible IRBs/IECs will be informed of any decisions made by the Sponsor based on recommendations from the DMC relating to subject safety that alter the conduct of this study. The Investigators will inform the subjects of such actions and the protocol, patient information sheet, and ICF will be revised, as appropriate.

## 13.9. Adjudication Committees

All suspected MACE, and drug-related hepatic injury events that occur after administration of the first dose of investigational product will be reviewed by the following blinded adjudication committees, depending on event type, before inclusion in any analysis. The 2 committees and event types they are responsible for adjudicating are as follows:

- Cardiovascular Adjudication Committee (CAC): Adjudicates all suspected MACE (Appendix D), including all deaths
- Hepatic Safety Committee: Adjudicates all suspected drug-related hepatic injury events

Each adjudication committee will have a charter that documents the reporting of events by the study site; definition of the suspected events to be adjudicated; supply of source documentation to the committee; and the entire data flow and process from committee membership, review of the events by the committee, reporting of the final assessment, and the working procedures of the committee.

The adjudication committee members will include experts with relevant adjudication experience; they will not be involved in the study as Investigators, DMC members, or consultants. Any candidate found to have a conflict or whose name is listed on the FDA debarment list will not be

offered membership. Conflicts of interest are assessed regularly, and if members are found to have a new conflict of interest they will be replaced.

The adjudication of suspected events will be based on available source documentation, including but not limited to individual clinical study data, hospital records, histology, discharge summaries, and/or death certificates. The adjudication committees will not receive any individual subject treatment or site-specific information. The assessment of events will be conducted in compliance with study-specific procedures, manuals, GCP, and all other applicable regulatory requirements, including the archiving of essential documents.

#### 14. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

### 14.1. Study Monitoring

Study records at each site will be monitored at regular intervals by a representative of the Sponsor, the CRA. The role of the CRA is to aid the Investigator in the maintenance and documentation of complete, accurate, legible, well organized and easily retrievable data. In addition, the CRA will ensure the Investigator's understanding of all applicable regulations concerning the clinical evaluation of the investigational product and will ensure an understanding of the protocol, reporting responsibilities and the validity of the data. This will include ensuring that full and appropriate essential documentation is available.

In order to perform this role, the CRA must perform source data verification and as such, must be given access to the subject's primary source documentation (eg, paper or electronic medical records such as consent to participate in the study, visit dates, screening and randomization numbers, demographic information, medical history, disease history, physical examination, vital signs, laboratory assessments [copy of laboratory reports], AEs, concomitant medications, dates of dispensing investigational product, ECGs, etc) that support data entries in the eCRF. The eCRF must be completed promptly after each visit to allow the progress and results of the study to be closely followed by the Medical Monitor.

The Investigator may exercise judgment in allowing the CRA access to particular sections of the subject's medical records if these are deemed irrelevant to the performance, observations or conduct of this study.

## 14.2. Audits and Inspections

The Investigator should understand that it may be necessary for the Sponsor, the IRB/IEC and/or a regulatory agency to conduct one or more site audits during or after the study and agrees to allow access to all study-related documentation and information and be available for discussion about the study.

## 15. QUALITY CONTROL AND QUALITY ASSURANCE

Logic and consistency checks will be performed on all data entered into the eCRF or ultimately transferred into the database to ensure accuracy and completeness.

Training sessions, regular monitoring of the study at the study site by the Sponsor or designated personnel (eg, CRA), instruction manuals, data verification, cross-checking and data audits will

be performed to ensure quality of all study data. Investigators' meetings and/or onsite study initiations will be performed to prepare Investigators and other study site personnel for appropriate collection of study data.

To ensure compliance with GCP and all applicable regulatory requirements, the Sponsor may conduct a quality assurance audit.

#### 16. ETHICS

#### 16.1. Ethics Review

The final study protocol, including the final version of the ICF and/or other subject information, must be approved or given a favorable opinion in writing by an IRB/IEC as appropriate. The Investigator must submit written IRB/IEC approval to the Sponsor before he or she can enroll any subject into the study. The Investigator is responsible for providing the IB and any other available safety information and information about payments and compensation available to study subjects to the ethics committee for review.

The Investigator is responsible for informing the IRB/IEC of any amendment to the protocol in accordance with local requirements. A favorable opinion on substantial amendments will be obtained prior to implementation, unless the amendment is necessary to reduce immediate risk to study participants. In addition, the IRB/IEC must approve all advertising used to recruit subjects for the study. The protocol must be reapproved by the IRB/IEC upon receipt of amendments and annually, as local regulations require.

The Investigator is also responsible for providing the IRB/IEC with reports of any reportable serious adverse drug reactions from any other study conducted with the investigational product. The Sponsor will provide this information to the Investigator.

Progress reports and notifications of SARs will be provided to the IRB/IEC according to local regulations and guidelines. Investigators or the Sponsor or its designee will provide reports to the IRB/IEC as requested, as a minimum annually, and after the study is complete.

## 16.2. Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/GCP, applicable regulatory requirements, and the Sponsor's policies.

#### 16.3. Written Informed Consent

The Investigator(s) at each center will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study. Subjects must also be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided.

The subject's signed and dated ICF must be obtained before conducting any study procedures.
The Investigator(s) must maintain the original, signed ICF. A copy of the ICF must be given to the subject.

#### 16.4. Subject Confidentiality and Data Protection

All information obtained during the conduct of the study with respect to the subject will be regarded as confidential and confidentiality of all subjects will be maintained. Monitors (eg, CRA, Medical Monitor), auditors and inspectors will require access to a subject's medical notes for the purpose of source document verification but the subject's confidentiality will be maintained at all times. An agreement for disclosure of any such information will be obtained in writing and is included in the statement of informed consent. The study data shall not be disclosed to a third party (with the exception of auditors and/or regulatory authorities) without the written consent of the Sponsor. All reports and communications relating to subjects in this study that are disclosed to an authorized third party will identify subjects only by protocol and assigned number and will be shared in a secure manner. All data shall be secured against unauthorized access.

The Investigator will maintain a list of subject names and identifying information (eg, subjects' hospital numbers, unique subject numbers). This list will not be collected by the Sponsor.

The written information sheet will explain that study data will be stored in a computer database, maintaining confidentiality in accordance with national data protection legislation. All data computer processed by the Sponsor or designee will be identified by unique subject number/randomization code/site number, only.

When personal subject data are stored or processed by computer, the data must be protected to prevent their disclosure to unauthorized third parties. The pertinent sections of the data protection laws in which the country is being conducted will be complied with in full.

The written information sheet and ICF will explain that, for data verification purposes, authorized representatives of the Sponsor, a regulatory authority, or an IRB/IEC may require direct access to parts of the hospital or study site records relevant to the study, including subject medical history.

#### 17. INVESTIGATOR OBLIGATIONS

The Investigator or a medically trained designee will be responsible for obtaining written informed consent and for the care of the subjects for the duration of the study. If the Investigator is not present at the study site during the assessment, he or she will leave instructions for the study site staff and a telephone number where he or she can be reached.

Named physician(s) will be responsible for the medical follow-up of subjects, as applicable.

#### 17.1. **AE Reporting**

The Investigator is responsible for recording AEs reported by the subject or discovered by any other means during the study. In agreeing to the provisions of this protocol, the Investigator accepts all legal responsibilities for immediate reporting of SAEs to the Sponsor.

#### 17.2. Protocol Deviations

The Investigator is not permitted to deviate from the protocol in any significant way without proper notification to the Sponsor (or designee). Only the Sponsor may amend the protocol. Any change in study conduct considered necessary by the Investigator will be made only after consultation with the Sponsor, who will then issue a formal protocol amendment to implement the change and obtain regulatory approval. The only exception is when the Investigator considers a subject's safety to be compromised if immediate action is not taken.

#### 17.3. Regulatory Documentation

The following regulatory documentation must be completed or provided, and maintained:

- Approved Patient Information Sheets and ICF (all versions)
- IRB/IEC approvals (of protocol/amendments, subject questionnaires, etc.)
- Form FDA 1572
- Current medical license of Principal Investigators
- Curriculum vitae of Principal Investigators
- Laboratory certification and reference ranges
- Financial disclosure forms

#### 17.4. Ethics Review

Please see Section 16.1 for the Investigator's responsibilities regarding ethics review.

#### 17.5. Archiving and Record Retention

The Investigator should retain all correspondence relating to this study in the Investigator Site File (ISF). Any study documents stored elsewhere should have their location referenced in the ISF.

All documents relating to the study including the ISF itself, source documents and subject medical files, completed study subject log and confidential subject identification list will be retained by the Investigator in accordance with regulations. US Federal regulations require that records of drug disposition, eCRFs, source documents, and all reports of this investigation shall be retained by the Investigator for a minimum of 2 years following notification by the Sponsor that the regulatory authorities have been notified of the study's termination, or 2 years following approval of the marketing application. If the Investigator is unable to retain the study documents for the required amount of time, the Sponsor must be notified of the individual who will be assuming this responsibility. In the event that storage of records becomes a problem at any time during this period, the Sponsor should be consulted for assistance. At the end of the minimum period, the Investigator should obtain written authorization from the Sponsor prior to the destruction of any records. The Investigator will notify the Sponsor if ownership of documents or responsibility for the study site is transferred. The Sponsor will inform Investigators should it become aware of any changes in storage requirements.

#### 18. PUBLICATION POLICY

The Sponsor intends to publish the results of all of the clinical studies that it Sponsors consistent with the Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013). Consistent with the recommendations of the editors of several leading medical journals, the International Committee of Medical Journal Editors (ICMJE), authorship of publications resulting from Intercept sponsored studies should fairly recognize the activities of those that have made a significant contribution to the study (http://www.icmje.org). Thus, it is anticipated that authorship will reflect the contribution made by the Sponsor personnel, the Investigators and others involved, such as statisticians.

In recent years, issues about conflicts of interest and accuracy of the study data have been raised in the medical press. Accordingly, the Sponsor has developed publication guidelines for clinical studies that are appropriate for this study. Key issues include the following:

- Clinical Study Registries (eg, clinicaltrials.gov): A description of the study and relevant design elements (eg, basic design, objectives and endpoints, sample size, study population, and key inclusion/exclusion criteria) and results (when available) will be published online in a manner consistent with applicable regulatory guidelines.
- Overview: Investigators, reviewers, and editors will have the right to audit the data to verify its accuracy.
- Responsibility: Each Investigator is responsible for the accuracy and completeness of all data from her/his site. The Sponsor (or its representatives) is responsible for the accuracy of the data entered into the study databases and the analyses conducted.
- Data Management: The Sponsor will establish data management and the SAP. The Investigators will have the opportunity to provide input into the plans. The Investigators will have the right to review the audit reports and data resolution decisions before the establishment of a clean file. The Investigators will have the right to appoint appropriately qualified auditors, with GCP experience, to audit the Sponsor's data before the establishment of a clean file. The Investigators must provide adequate notice (at least 2 months) to the Sponsor of their intention to audit a study. The audit should be conducted in a timely manner to allow the resolution of discrepancies before a clean file is established. The Investigators will bear all the costs for the conduct of audits that they initiate, except those related to the resolution of data queries which the Sponsor will bear. Such audits must be conducted in such a manner as to minimize the time to create the clean file.
- Authorship: The Sponsor, in collaboration with the Investigators, will establish the appropriate authorship and responsibility for drafting study documents in accordance with the principles of the ICMJE. All manuscripts will be reviewed and agreed upon before submission for publication by all authors.
- Single Center Publication and Additional Publications: This is a multicenter study and is designed to be published with complete data from all the study sites. Single center publications are therefore not considered appropriate. Any such publications should clearly state that the data are "extracted" from a multicenter study and that the

study was not intended, or statistically powered, for data presentation by a single study site.

- Intercept Review of External Manuscripts: Consistent with this, Investigators must submit any drafts of any publications or presentations that may arise from this study to the Sponsor for review and approval and to ensure consistency with the policy in this protocol at least 30 days before submission for publication or presentation. The Sponsor will have the right to request appropriate modification to correct facts and to represent its, or the Publication Committee's, opinion if these differ with the proposed publication.
- Confidentiality: Investigators will conduct all interactions with the company and
  with third parties consistent with the executed confidentiality agreements. While
  publication, by intention, presents the critical scientific data in a public forum, some
  information (such as future plans, results of preclinical studies, or chemical formulae)
  may still need to remain confidential.
- Medical Journal Review: Upon request, all pertinent study data and information will be made available as supplemental information for journal editors and reviewers to evaluate and audit (eg, protocol and amendments, data tabulations, etc).
   Arrangements will be made to maintain the confidentiality of such supplemental information. Arrangements will also be made to maintain the confidentiality of the identity of journal reviewers. Records will be maintained of which documents and datasets were reviewed.

#### 19. LIST OF REFERENCES

Adorini L, Pruzanski M, Shapiro D. Farnesoid X receptor targeting to treat nonalcoholic steatohepatitis. Drug Discov Today. 2012 Sep;17(17-18):988-997.

Albanis E, Alvarez CE, Pruzanski M, et al. INT-747, a novel FXR activator, reverses hepatic fibrosis and cirrhosis in thiocetamideinduced liver injury in rats. Hepatology. 2005;42(Supplement 1):Abstract 1040.

American Diabetes Association. Standards of medical care in diabetes-2013. Diabetes Care. 2013;36(Suppl 1):S11-S66.

Angulo P. Clinical trials: Trial design in NASH–realities and challenges. NatRev. Gastroenterol Hepatol. 2011 Aug;8(8):424-425.

Athyros VG, Tziomalos K, Gossios TD, et al. Safety and efficacy of long-term statin treatment for cardiovascular events in patients with coronary heart disease and abnormal liver tests in the Greek Atorvastatin and Coronary Heart Disease Evaluation (GREACE) Study: a post-hoc analysis. Lancet. 2010 Dec 4;376(9756):1916-1922.

Belfort R, Harrison SA, Brown K, et al. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-2307.

Beuers U, Gershwin ME, Gish RG, et al. Changing nomenclature for PBC: From 'cirrhosis' to 'cholangitis'. Dig Liver Dis. 2015a;47(11):924-6.

Beuers U, Gershwin ME, Gish RG, et al. Changing nomenclature for PBC: From 'cirrhosis' to 'cholangitis'. Gastroenterology. 2015b;149(6):1627-9.

Beuers U, Gershwin ME, Gish RG, et al. Changing nomenclature for PBC: From 'cirrhosis' to 'cholangitis'. Hepatology. 2015c;62(5):1620-2.

Calderon RM, Cubeddu LX, Goldberg RB, et al. Statins in the treatment of dyslipidemia in the presence of elevated liver aminotransferase levels: a therapeutic dilemma. Mayo Clinic proceedings. 2010 Apr;85(4):349-356.

Cariou B, van Harmelen K, Duran-Sandoval D, et al. The farnesoid X receptor modulates adiposity and peripheral insulin sensitivity in mice. J Biol Chem. 2006 Apr 21;281(16):11039-11049.

CEREP. In Vitro pharmacology:High-throughput profile - Study of INT-747. 2008 June 7, 2008;Study #14862.

Chalasani N, Younossi Z, Lavine JE, et al. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-2023.

Cromwell WC, Otvos JD, Keyes MJ, et al. LDL Particle Number and Risk of Future Cardiovascular Disease in the Framingham Offspring Study - Implications for LDL Management. J Clin Lipidol. 2007 Dec;1(6):583-592.

Desai CS, Martin SS, Blumenthal RS. Non-cardiovascular effects associated with statins. BMJ 2014;349:g3743.

Ekstedt M, Hagstrom H, Nasr P, et al. Fibrosis stage is the strongest predictor for disease-specific mortality in NAFLD after up to 33 years of follow-up. Hepatology. 2015;61:1547-1554.

Ertle J, Dechene A, Sowa JP, et al. Non-alcoholic fatty liver disease progresses to hepatocellular carcinoma in the absence of apparent cirrhosis. Int J Cancer. 2011 May 15;128(10):2436-2443.

FDA. Guidance for Industry Drug-Induced Liver Injury:Premarketing Clinical Evaluation. Drug Safety Report. 2009 July.

Fu L, John LM, Adams SH, et al. Fibroblast growth factor 19 increases metabolic rate and reverses dietary and leptin-deficient diabetes. Endocrinology. 2004 Jun;145(6):2594-2603.

Gadaleta RM, van Erpecum KJ, Oldenburg B, et al. Farnesoid X receptor activation inhibits inflammation and preserves the intestinal barrier in inflammatory bowel disease. Gut. 2011 Apr;60(4):463-472.

Gautier T, de Haan W, Grober J, et al. Farnesoid X receptor activation increases cholesteryl ester transfer protein expression in humans and transgenic mice. J Lipid Res. 2013 Aug;54(8):2195-2205.

Hartman HB, Gardell SJ, Petucci CJ, et al. Activation of farnesoid X receptor prevents atherosclerotic lesion formation in LDLR-/- and apoE-/- mice. J Lipid Res. 2009 Jun;50(6):1090-1100.

Jackevicius CA, Chou MM, Ross JS, et al. Generic atorvastatin and health care costs. N Engl J Med. 2012 Jan 19;366(3):201-204.

Jackevicius CA, Tu JV, Krumholz HM. Statins: is it safe and effective to use generic "equivalents"? Can J Cardiol. 2013 Apr;29(4):408-410.

Jeyarajah EJ, Cromwell WC, Otvos JD. Lipoprotein particle analysis by nuclear magnetic resonance spectroscopy. Clin Lab Med. 2006 Dec;26(4):847-870.

Kleiner D, Brunt E, Van Natta M, et al. Design and Validation of a Histological Scoring System for Nonalcoholic Fatty Liver Disease. Hepatology. 2005;41:1313-1321.

Lefebvre P, Cariou B, Lien F, et al. Role of bile acids and bile acid receptors in metabolic regulation. Physiol Rev. 2009 Jan;89(1):147-191.

Li YT, Swales KE, Thomas GJ, et al. Farnesoid x receptor ligands inhibit vascular smooth muscle cell inflammation and migration. Arterioscler Thromb Vasc Biol. 2007 Dec;27(12):2606-2611.

Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-690.

Ma K, Saha PK, Chan L, et al. Farnesoid X receptor is essential for normal glucose homeostasis. J Clin Invest. 2006 Apr;116(4):1102-1109.

Mampuya WM, Frid D, Rocco M, et al. Treatment strategies in patients with statin intolerance: the Cleveland Clinic experience. Am Heart J. 2013;166:597-603.

McGowan MP, Treating to New Target Study G. There is no evidence for an increase in acute coronary syndromes after short-term abrupt discontinuation of statins in stable cardiac patients. Circulation. 2004 Oct 19;110(16):2333-2335.

Mencarelli A, Renga B, Distrutti E, et al. Antiatherosclerotic effect of farnesoid X receptor. American journal of physiology Heart and circulatory physiology. 2009 Feb;296(2):H272-H281.

Miyazaki-Anzai S, Levi M, Kratzer A, et al. Farnesoid X receptor activation prevents the development of vascular calcification in ApoE-/- mice with chronic kidney disease. Circ Res. 2010 Jun 25;106(12):1807-1817.

Mookerjee RP, Mehta G, Balasubramaniyan V, et al. Hepatic dimethylarginine-dimethylaminohydrolase1 is reduced in cirrhosis and is a target for therapy in portal hypertension. J Hepatol. 2015;62:325-331.

Mudaliar S, Henry RR, Sanyal AJ, et al. Efficacy and safety of the farnesoid X receptor agonist obeticholic acid in patients with type 2 diabetes and nonalcoholic fatty liver disease. Gastroenterology. 2013 Sep;145(3):574-582 e1.

Neuschwander-Tetri BA, Brunt EM, Wehmeier KR, et al. Improved nonalcoholic steatohepatitis after 48 weeks of treatment with the PPAR-gamma ligand rosiglitazone. Hepatology. 2003 Oct;38(4):1008-1017.

Neuschwander-Tetri BA, Loomba R, Sanyal AJ, et al. Farnesoid X nuclear receptor ligand obeticholic acid for non-cirrhotic, non-alcoholic steatohepatitis (FLINT): a multicentre, randomised, placebo-controlled trial. The Lancet. 2014;S0140-6736:1-11.

NICE. Lipid Modification: Cardiovascular Risk Assessment and the Modification of Blood Lipids for the Primary and Secondary Prevention of Cardiovascular Disease. National Institute for Health and Clinical Excellence: Guidance. London 2014.

Nissen SE, Tardif JC, Nicholls SJ, et al. Effect of torcetrapib on the progression of coronary atherosclerosis. N Engl J Med. 2007 Mar 29;356(13):1304-1316.

Organisation WG. World Gastroenterology Organisation Global Guidelines: nonalcoholic fatty liver disease and nonalcholic steatohepatitis. 2012 June.

Otvos JD, Collins D, Freedman DS, et al. Low-density lipoprotein and high-density lipoprotein particle subclasses predict coronary events and are favorably changed by gemfibrozil therapy in the Veterans Affairs High-Density Lipoprotein Intervention Trial. Circulation. 2006 Mar 28;113(12):1556-1563.

Pagadala MR, McCullough AJ. The relevance of liver histology to predicting clinically meaningful outcomes in nonalcoholic steatohepatitis. Clin Liver Dis. 2012 Aug;16(3):487-504.

Pastori D, Polimeni L, Baratta F, et al. The efficacy and safety of statins for the treatment of non-alcoholic fatty liver disease. Digestive and liver disease: official journal of the Italian Society of Gastroenterology and the Italian Association for the Study of the Liver. 2015 Jan;47(1):4-11.

Pellicciari R, Fiorucci S, Camaioni E, et al. 6alpha-ethyl-chenodeoxycholic acid (6-ECDCA), a potent and selective FXR agonist endowed with anticholestatic activity. J Med Chem. 2002 Aug 15;45(17):3569-3572.

Perk J, De Backer G, Gohlke H, et al. European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-1701.

Rizzo G, Disante M, Mencarelli A, et al. The farnesoid X receptor promotes adipocyte differentiation and regulates adipose cell function in vivo. Mol Pharmacol. 2006 Oct;70(4):1164-1173.

Rizzo G, Passeri D, De Franco F. In vitro human ERG inhibition by INT-747. Internal Report hERG-001. 2009.

Rohatgi A, Khera A, Berry JD, et al. HDL Cholesterol Efflux Capacity and Incident Cardiovascular Events. N Engl J Med. 2014 Dec 18;371(25):2383-2393.

Rosenson RS, Baker SK, Jacobson TA et al. An assessment by the statin muscle safety task force: 2014 update. J Clin Lipid. 2014;8:S58-S71.

Sanyal AJ, Chalasani N, Kowdley KV, et al. Pioglitazone, vitamin E, or placebo for nonalcoholic steatohepatitis. N Engl J Med. 2010 May 6;362(18):1675-1685.

Saunders JB, Aasland OG, Babor TF. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804.

Savkur RS, Thomas JS, Bramlett KS, et al. Ligand-dependent coactivation of the human bile acid receptor FXR by the peroxisome proliferator-activated receptor gamma coactivator-1alpha. J Pharmacol Exp Ther. 2005 Jan;312(1):170-178.

Shulman AI, Mangelsdorf DJ. Retinoid x receptor heterodimers in the metabolic syndrome. N Engl J Med. 2005 Aug 11;353(6):604-615.

Simic I, Reiner Z. Adverse effects of statins – myths and reality. Curr Pharm Des. 2015;21:1220-1226.

Stone NJ, Robinson JG, Lichtenstein AH, et al. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-2934.

Teramoto T, Sawada T, Iwamoto K, et al. Clinical efficacy and tolerability of ezetimibe in combination with atorvastatin in Japanese patients with hypercholesterolemia-ezetimibe phase IV randomized controlled trial in patients with hypercholesterolemia. Curr Ther Res Clin Exp. 2012 Feb;73(1-2):16-40.

Teramoto T, Takeuchi M, Morisaki Y, et al. Efficacy, safety, tolerability, and pharmacokinetic profile of evacetrapib administered as monotherapy or in combination with atorvastatin in Japanese patients with dyslipidemia. Am J Cardiol. 2014 Jun 15;113(12):2021-2029.

Tikkanen MJ, Fayyad R, Faergeman O, et al. Effect of intensive lipid lowering with atorvastatin on cardiovascular outcomes in coronary heart disease patients with mild-to-moderate baseline elevations in alanine aminotransferase levels. Int J Cardiol. 2013 Oct 9;168(4):3846-3852.

Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-285.

Wang XX, Jiang T, Shen Y, et al. The farnesoid X receptor modulates renal lipid metabolism and diet-induced renal inflammation, fibrosis, and proteinuria. Am J Physiol Renal Physiol. 2009 Dec;297(6):F1587-F1596.

Wang XX, Jiang T, Shen Y, et al. Diabetic nephropathy is accelerated by farnesoid X receptor deficiency and inhibited by farnesoid X receptor activation in a type 1 diabetes model. Diabetes. 2010 Nov;59(11):2916-2927.

Wang YD, Chen WD, Wang M, et al. Farnesoid X receptor antagonizes nuclear factor kappaB in hepatic inflammatory response. Hepatology. 2008 Nov;48(5):1632-1643.

Watanabe M, Houten SM, Wang L, et al. Bile acids lower triglyceride levels via a pathway involving FXR, SHP, and SREBP-1c. J Clin Invest. 2004 May;113(10):1408-1418.

Williams R, Horton R. Liver disease in the UK: a Lancet Commission. Lancet. 2013 Nov 9:382(9904):1537-1538.

Xu J, Stanislaus S, Chinookoswong N, et al. Acute glucose-lowering and insulin-sensitizing action of FGF21 in insulin-resistant mouse models--association with liver and adipose tissue effects. Am J Physiol Endocrinol Metab. 2009 Nov;297(5):E1105-E1114.

Younossi ZM, Stepanova M, Rafiq N, et al. Pathologic criteria for nonalcoholic steatohepatitis: interprotocol agreement and ability to predict liver-related mortality. Hepatology. 2011 Jun;53(6):1874-1882.

Zhang H, Plutzky J, Skentzos S, et al. Discontinuation of statins in routine care settings: a cohort study. Ann Intern Med. 2013:158:526-534.

Zhang S, Wang J, Liu Q, et al. Farnesoid X receptor agonist WAY-362450 attenuates liver inflammation and fibrosis in murine model of non-alcoholic steatohepatitis. J Hepatol. 2009 Aug;51(2):380-388.

Zhang Y, Lee FY, Barrera G, et al. Activation of the nuclear receptor FXR improves hyperglycemia and hyperlipidemia in diabetic mice. Proc Natl Acad Sci U S A. 2006 Jan 24;103(4):1006-1011.

Zhang Y, Edwards PA. FXR signaling in metabolic disease. FEBS Lett. 2008 Jan 9;582(1):10-18.

Zhang Y, Yin L, Anderson J, et al. Identification of novel pathways that control farnesoid X receptor-mediated hypocholesterolemia. J Biol Chem. 2010 Jan 29;285(5):3035-3043.

## APPENDIX A. AMERICAN COLLEGE OF CARDIOLOGY/AMERICAN HEART ASSOCIATION GUIDANCE FOR THE USE OF STATINS

#### **PRACTICE GUIDELINE**

# **2013 ACC/AHA Guideline on the Treatment of Blood Cholesterol to Reduce Atherosclerotic Cardiovascular Risk in Adults**



A Report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines

Endorsed by the American Academy of Physician Assistants, American Association of Cardiovascular and Pulmonary Rehabilitation, American Pharmacists Association, American Society for Preventive Cardiology, Association of Black Cardiologists, Preventive Cardiovascular Nurses Association, and WomenHeart: The National Coalition for Women With Heart Disease

### Expert Panel Members

Neil J. Stone, MD, MACP, FAHA, FACC, Chair

Jennifer G. Robinson, MD, MPH, FAHA, Vice Chair

Alice H. Lichtenstein, DSc, FAHA, Vice Chair

C. Noel Bairey Merz, MD, FAHA, FACC Conrad B. Blum, MD, FAHA Robert H. Eckel, MD, FAHA Anne C. Goldberg, MD, FACP, FAHA

David Gordon, MD\*

Methodology Members Karen M. Eddleman, BS Nicole M. Jarrett Ken LaBresh, MD Daniel Levy, MD\*

Donald M. Lloyd-Jones, MD, ScM, FACC, FAHA

Patrick McBride, MD, MPH, FAHA

J. Sanford Schwartz, MD

Susan T. Shero, MS, RN\*

Sidney C. Smith, JR, MD, FACC, FAHA Karol Watson, MD, PhD, FACC, FAHA

Peter W. F. Wilson, MD, FAHA

\*Ex-Officio Members.

Lev Nevo, MD Janusz Wnek, PHD

#### ACC/AHA Task Force Members

**Guidelines** 

Jeffrey L. Anderson, MD, FACC, FAHA, *Chair* Jonathan L. Halperin, MD, FACC, FAHA, *Chair-Elect* 

Nancy M. Albert, PhD, CCNS, CCRN, FAHA Biykem Bozkurt, MD, PhD, FACC, FAHA Ralph G. Brindis, MD, MPH, MACC Lesley H. Curtis, PhD, FAHA

**Subcommittee on** Sidney C. Smith, JR, MD, FACC, FAHA, *Chair* **Prevention** 

David DeMets, PHD

Judith S. Hochman, MD, FACC, FAHA Richard J. Kovacs, MD, FACC, FAHA E. Magnus Ohman, MD, FACC Susan J. Pressler, PhD, RN, FAAN, FAHA Frank W. Sellke, MD, FACC, FAHA Win-Kuang Shen, MD, FACC, FAHA

Gordon F. Tomaselli, MD, FACC, FAHA, Co-Chair

The American College of Cardiology requests that this document be cited as follows: Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PWF. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol 2014;63:2889–934.

This article is copublished in Circulation.

Copies: This document is available on the World Wide Web sites of the American College of Cardiology (http://www.cardiosource.org) and the American Heart Association (my.americanheart.org). For copies of this document, please contact the Elsevier Inc. Reprint Department, fax (212) 462-1935, e-mail reprints@elsevier.com.

The Journal of the American College of Cardiology is published on behalf of the American College of Cardiology Foundation by Elsevier Inc.; Circulation is published on behalf of the American Heart Association, Inc., by Wolters Kluwer. This is an open access article under the terms of the Creative Commons Attribution Non-Commercial-NoDervis License, which permits use, distribution, and reproduction in any medium, provided that the Contribution is properly cited, the use is noncommercial, and no modifications or adaptations

are made.

This document was approved by the American College of Cardiology Board of Trustees and the American Heart Association Science Advisory and Coordinating Committee in November 2013. The Academy of Nutrition and Dietetics affirms the value of this guideline.

| T. | ABLE | OF CONTENTS |
|---|---|---|
| | | e and Transition to ACC/AHA Guidelines to<br>Cardiovascular Risk2890 |
| 1. | Intro | <b>oduction</b> |
| | 1.1. | Organization of the Panel |
| | | Document Review and Approval 2891 |
| | 1.3. | <b>Scope of Guideline</b> |
| | 1.4. | Methodology and Evidence Review 2894 |
| 2. | Ove | rview of the Guideline2895 |
| | 2.1. | Lifestyle as the Foundation for |
| | 2.2 | ASCVD Risk-Reduction Efforts |
| 3. | | Initiation of Statin Therapy |
| <b>3.</b> | Criti | cai Questions and Conclusions2897 |
| | 3.1. | Identification of CQs |
| | | 3.1.1. CQ1: LDL-C and Non-HDL-C Goals in |
| | | Secondary Prevention |
| | | Primary Prevention |
| | | 3.1.3. CQ3: Efficacy and Safety of |
| | | Cholesterol-Lowering Medications 2899 |
| 4. | Stat | in Treatment: Recommendations2899 |
| | 4.1. | Intensity of Statin Therapy in Primary and |
| | | Secondary Prevention |
| | 4.2. | LDL-C and Non-HDL-C Treatment Goals $\dots 2901$ |
| | 4.3. | Secondary Prevention |
| | 4.4. | Primary Prevention in Individuals ≥21 Years of Age With LDL-C ≥190 mg/dL |
| | 4.5 | Primary Prevention in Individuals With |
| | 1101 | <b>Diabetes</b> |
| | 4.6. | Primary Prevention in Individuals Without |
| | | Diabetes and With LDL-C 70 to 189 mg/dL 2905 |
| | 4.7. | Risk Assessment in Primary Prevention 2906 |
| | 4.8. | Heart Failure and Hemodialysis |
| 5. | Safe | ety: Recommendations |
| 6. | Man | aging Statin Therapy: |
| • | | ommendations |
| | 6.1. | Monitoring Statin Therapy |
| | | Optimizing Statin Therapy |
| | | Insufficient Response to Statin Therapy 2912 |
| | | 6.3.1. Testing |
| _ | | Statin-Intolerant Individuals 2913 |
| 7. | | ected Clinical and Population groups2913 |
| | 7.1. | Sex and Racial and Ethnic Subgroups 2913 |
| | | Individuals >75 Years of Age |

| 8. | <b>Limitations</b> |
|-----|-----------------------------------------------------------------------|
| 9. | Evidence Gaps and Future Research Needs2914 |
| 10. | Conclusions |
| Ref | erences |
| | endix 1. Author Relationships With Industry Other Entities (Relevant) |
| | endix 2. Expert Reviewer Relationships With ustry and Other Entities |
| App | endix 3. Abbreviations2923 |
| Арр | endix 4. Evidence Statements2923 |
| | endix 5. Expanded Discussion of at's New in the Guideline |

### Preamble and Transition to ACC/AHA Guidelines to Reduce Cardiovascular Risk

The goals of the American College of Cardiology (ACC) and the American Heart Association (AHA) are to prevent cardiovascular diseases; improve the management of people who have these diseases through professional education and research; and develop guidelines, standards, and policies that promote optimal patient care and cardiovascular health. Toward these objectives, the ACC and AHA have collaborated with the National Heart, Lung, and Blood Institute (NHLBI) and stakeholder and professional organizations to develop clinical practice guidelines for assessment of cardiovascular risk, lifestyle modifications to reduce cardiovascular risk, management of blood cholesterol in adults, and management of overweight and obesity in adults.

In 2008, the NHLBI initiated these guidelines by sponsoring rigorous systematic evidence reviews for each topic by expert panels convened to develop critical questions (CQs), interpret the evidence, and craft recommendations. In response to the 2011 report from the Institute of Medicine on the development of trustworthy clinical guidelines (1), the NHLBI Advisory Council recommended that the NHLBI focus specifically on reviewing the highest-quality evidence and partner with other organizations to develop recommendations (2,3). Accordingly, in June 2013 the NHLBI initiated collaboration with the ACC and AHA to work with other organizations to complete and publish the 4 guidelines noted above and make them available to the widest possible constituency. Recognizing that the Expert Panels/Work Groups did not

consider evidence beyond 2011 (except as specified in the methodology), the ACC, AHA, and collaborating societies plan to begin updating these guidelines starting in 2014.

The joint ACC/AHA Task Force on Practice Guide-lines (Task Force) appointed a subcommittee to shepherd this transition, communicate the rationale and expectations to the writing panels and partnering organizations, and expeditiously publish the documents. The ACC/AHA and partner organizations recruited a limited number of expert reviewers for fiduciary examination of content, recognizing that each document had undergone extensive peer review by representatives of the NHLBI Advisory Council, key federal agencies, and scientific experts. Each writing panel responded to comments from these reviewers. Clarifications were incorporated where appropriate, but there were no substantive changes because the bulk of the content was undisputed.

Although the Task Force led the final development of these prevention guidelines, they differ from other ACC/ AHA guidelines. First, as opposed to an extensive compendium of clinical information, these documents are significantly more limited in scope and focus on selected CQs on each topic, based on the highest-quality evidence available. Recommendations were derived from randomized trials, meta-analyses, and observational studies evaluated for quality and were not formulated when sufficient evidence was not available. Second, the text accompanying each recommendation is succinct, summarizing the evidence for each question. The Full Panel/Work Group Reports include more detailed information about the evidence statements that serve as the basis for recommendations. Third, the format of the recommendations differs from other ACC/ AHA guidelines. Each recommendation has been mapped from the NHLBI grading format to the ACC/AHA Classification of Recommendation/Level of Evidence (COR/ LOE) construct (Table 1) and is expressed in both formats. Because of the inherent differences in grading systems and the clinical questions driving the recommendations, alignment between the NHLBI and ACC/AHA formats is in some cases imperfect. Explanations of these variations are noted in the recommendation tables, where applicable.

In consultation with NHLBI, the policies adopted by the writing panels to manage relationships of authors with industry and other entities (RWI) are outlined in the methods section of each panel report. These policies were in effect when this effort began in 2008 and throughout the writing process and voting on recommendations, until the process was transferred to ACC/AHA in 2013. In the interest of transparency, the ACC/AHA requested that panel authors resubmit RWI disclosures as of July 2013. Relationships relevant to this guideline are disclosed in Appendix 1. None of the ACC/AHA expert reviewers had relevant RWI (Appendix 2). See Appendix 3 for a list of abbreviations used in the guideline.

Systematic evidence reports and accompanying summary tables were developed by the expert panels and

NHLBI. The guideline was reviewed by the ACC/AHA Task Force and approved by the ACC Board of Trustees, and the AHA Science Advisory and Coordinating Committee. In addition, ACC/AHA sought endorsement from other stakeholders, including professional organizations. It is the hope of the writing panels, stakeholders, professional organizations, NHLBI, and Task Force that the guidelines will garner the widest possible readership for the benefit of patients, providers, and the public health.

These guidelines are meant to define practices that meet the needs of patients in most circumstances and are not a replacement for clinical judgment. The ultimate decision about care of a particular patient must be made by the healthcare provider and patient in light of the circumstances presented by that patient. As a result, situations might arise in which deviations from these guidelines may be appropriate. These considerations notwithstanding, in caring for most patients, clinicians can employ the recommendations confidently to reduce the risks of atherosclerotic cardiovascular disease (ASCVD) events.

See Tables 1a and 1b for an explanation of the NHLBI recommendation grading methodology.

#### 1. Introduction

#### 1.1. Organization of the Panel

The Blood Cholesterol Expert Panel (Expert Panel) was originally convened as the Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel IV) appointed by the NHLBI. The Expert Panel was composed of 13 members and 3 ex-officio members, which included primary care physicians, cardiologists, endocrinologists, and experts in clinical lipidology, clinical trials, cardiovascular epidemiology and nutrition, and guideline development. The Expert Panel chair asked all panel members to disclose any conflict-of-interest information to the full panel in advance of the deliberations; members with conflicts were asked to recuse themselves from voting on any aspect of the guideline for which a conflict might exist. All 16 members of the NHLBI Adult Treatment Panel IV Panel transitioned to the ACC/AHA guideline Expert Panel. Independent contractors performed the systematic review with the assistance of the Expert Panel and provided methodological guidance to the Expert Panel.

#### 1.2. Document Review and Approval

A formal peer review process was initially completed under the auspices of the NHLBI and included 23 expert reviewers and representatives of federal agencies. This document was also reviewed by 4 expert reviewers nominated by the ACC and the AHA when the management of the guideline transitioned to the ACC/AHA. The ACC and

Table 1. Applying Classification of Recommendation and Level of Evidence

| | | SIZE OF TREA | TMENT EFFECT | |
|---|---|---|---|---|
| | CLASS I Benefit >>> Risk Procedure/Treatment SHOULD be performed/ administered | CLASS IIa Benefit >> Risk Additional studies with focused objectives needed IT IS REASONABLE to perform procedure/administer treatment | CLASS IIb Benefit ≥ Risk Additional studies with broad objectives needed; additional registry data would be helpful Procedure/Treatment MAY BE CONSIDERED | CLASS III No Benefit or CLASS III Harm Procedure/ Test Treatment COR III: Not No Proven No benefit Helpful Benefit COR III: Excess Cost Harmful W/O Benefit to Patients or Harmful |
| LEVEL A Multiple populations evaluated* Data derived from multi randomized clinical trial or meta-analyses LEVEL B Limited populations evaluated* Data derived from a single randomized trial or nonrandomized studi LEVEL C Very limited populations evaluated* Only consensus opinion of experts, case studies or standard of care | IIIUILIDIE TAIIUUIIIIZEU LITAIS | ■ Recommendation in favor of treatment or procedure being useful/effective ■ Some conflicting evidence from multiple randomized trials or meta-analyses | ■ Recommendation's usefulness/efficacy less well established ■ Greater conflicting evidence from multiple randomized trials or meta-analyses | ■ Recommendation that procedure or treatment is not useful/effective and may be harmful ■ Sufficient evidence from multiple randomized trials or meta-analyses |
| LEVEL B Limited populations evaluated* Data derived from a single randomized trial or nonrandomized studi | ■ Recommendation that procedure or treatment is useful/effective ■ Evidence from single randomized trial or nonrandomized studies | ■ Recommendation in favor of treatment or procedure being useful/effective ■ Some conflicting evidence from single randomized trial or nonrandomized studies | ■ Recommendation's usefulness/efficacy less well established ■ Greater conflicting evidence from single randomized trial or nonrandomized studies | ■ Recommendation that procedure or treatment is not useful/effective and may be harmful ■ Evidence from single randomized trial or nonrandomized studies |
| LEVEL C Very limited populations evaluated* Only consensus opinion of experts, case studies or standard of care | useful/effective Only expert opinion, case studies or standard of care | ■ Recommendation in favor of treatment or procedure being useful/effective ■ Only diverging expert opinion, case studies, or standard of care | ■ Recommendation's usefulness/efficacy less well established ■ Only diverging expert opinion, case studies, or standard of care | ■ Recommendation that procedure or treatment is not useful/effective and may be harmful ■ Only expert opinion, case studies, or standard of care |
| Suggested phrases for writing recommendations | should<br>is recommended<br>is indicated<br>is useful/effective/beneficial | is reasonable<br>can be useful/effective/beneficial<br>is probably recommended<br>or indicated | may/might be considered<br>may/might be reasonable<br>usefulness/effectiveness is<br>unknown/unclear/uncertain<br>or not well established | COR III: COR III: No Benefit Harm is not potentially recommended harmful is not indicated causes harm should not be associated with |
| Comparative<br>effectiveness phrases <sup>†</sup> | treatment/strategy A is recommended/indicated in preference to treatment B treatment A should be chosen over treatment B | treatment/strategy A is probably recommended/indicated in preference to treatment B it is reasonable to choose treatment A over treatment B | | performed/ excess morbid-<br>administered/ ity/mortality<br>other should not be<br>is not useful/ performed/<br>beneficial/ administered/<br>effective other |

A recommendation with Level of Evidence B or C does not imply that the recommendation is weak. Many important clinical questions addressed in the guidelines do not lend themselves to clinical trials. Even when randomized trials are unavailable, there may be a very clear clinical consensus that a particular test or therapy is useful or effective.

AHA reviewers' RWI information is published in this document (Appendix 2).

This document was approved for publication by the governing bodies of the ACC and AHA and endorsed by the American Academy of Physician Assistants, American Association of Cardiovascular and Pulmonary Rehabilitation, American Pharmacists Association, American Society for Preventive Cardiology, Association of Black Cardiologists, Preventive Cardiovascular Nurses Association, and WomenHeart: The National Coalition for Women with Heart Disease.

#### 1.3. Scope of Guideline

This guideline is based on the Full Panel Report, which is provided as an online-only data supplement to the

guideline. The Full Panel Report contains background and additional material related to content, methodology, evidence synthesis, rationale, and references and is supported by the NHLBI Systematic Evidence Review, which can be found at http://www.nhlbi.nih.gov/guidelines/cholesterol/ser/. Table 2 provides an overview to facilitate understanding what is new in the present guideline.

The Expert Panel was charged with using data from randomized controlled trials (RCTs) and systematic reviews and meta-analyses of RCTs to update the clinical practice recommendations for the treatment of blood cholesterol levels to reduce ASCVD risk. For this guideline, ASCVD includes coronary heart disease (CHD), stroke, and peripheral arterial disease, all of presumed atherosclerotic origin. These recommendations are intended to provide a

<sup>\*</sup>Data available from clinical trials or registries about the usefulness/efficacy in different subpopulations, such as sex, age, history of diabetes, history of prior myocardial infarction, history of heart failure, and prior aspirin use.

<sup>†</sup>For comparative-effectiveness recommendations (Class I and IIa; Level of Evidence A and B only), studies that support the use of comparator verbs should involve direct comparisons of the treatments or strategies being evaluated.

Grade

| rabie 1a. | MHLBI | Grading | OT | tne | Strengtn | 01 |
|-----------|---------|---------|----|-----|----------|----|
| Recomme | ndation | S | | | | |

#### Strong recommendation

There is high certainty based on evidence that the net benefit is substantial.

#### Moderate recommendation

There is moderate certainty based on evidence that the net benefit is moderate to substantial, or there is high certainty that the net benefit is moderate.

Strength of Recommendation\*

#### Weak recommendation

There is at least moderate certainty based on evidence that there is a small net benefit.

#### Recommendation against

There is at least moderate certainty based on evidence that there is no net benefit or that risks/harms outweigh benefits.

#### Expert opinion ("There is insufficient evidence or evidence is unclear or conflicting, but this is what the Work Group recommends.")

Net benefit is unclear. Balance of benefits and harms cannot be determined because of no evidence, insufficient evidence, unclear evidence, or conflicting evidence, but the Work Group thought it was important to provide clinical guidance and make a recommendation. Further research is recommended in this area.

#### No recommendation for or against ("There is insufficient evidence or evidence is unclear or conflicting.")

Net benefit is unclear. Balance of benefits and harms cannot be determined because of no evidence, insufficient evidence, unclear evidence, or conflicting evidence, and the Work Group thought no recommendation should be made. Further research is recommended in this area.

†Net benefit is defined as benefits minus risks/harms of the service/intervention. ECG indicates electrocardiogram; MI, myocardial infarction; and NHLBI, National Heart, Lung, and Blood Institute.

strong, evidence-based foundation for the treatment of cholesterol for the primary and secondary prevention of ASCVD in women and men.

Because RCT data were used to identify those *most likely* to benefit from cholesterol-lowering statin therapy, the recommendations will be of value to primary care clinicians as well as specialists concerned with ASCVD prevention. Importantly, the recommendations were designed to be easy to use in the clinical setting, facilitating the implementation of a strategy of risk assessment and treatment focused on the prevention of ASCVD. The present guideline is intended to address treatment of adults (≥21 years of age) to complement the NHLBI cardiovascular health risk-reduction guideline for children and adoles-

The members of the Expert Panel acknowledge the important contributions arising from decades of genetic and biochemical studies, observational epidemiological and ecological studies, and in vitro and animal experiments that associated higher low-density lipoprotein

Table 1b. NHLBI Quality Rating of the Strength of Evidence

| Type of Evidence | Quality Rating* |
|---|---|
| well-designed, well-executed† RCT that adequately represent populations to which the results are applied and directly assess effects on health outcomes. Meta-analyses of such studies. Highly certain about the estimate of effect. Further esearch is unlikely to change our confidence in the estimate of effect. | High |
| o RCT with minor limitations‡ affecting confidence in, or applicability of, the results. O Well-designed, well-executed nonrandomized controlled studies§ and well-designed, well-executed observational studies . O Meta-analyses of such studies. Moderately certain about the estimate of effect. Further esearch may have an impact on our confidence in the estimate of effect and may change the estimate. | Moderate |
| PRCT with major limitations. Nonrandomized controlled studies and observational studies with major limitations affecting confidence in, or applicability of, the results. Uncontrolled clinical observations without an appropriate comparison group (e.g., case series, case reports). Physiological studies in humans. Meta-analyses of such studies. Ow certainty about the estimate of effect. Further esearch is likely to have an impact on our confidence in the estimate of effect and is likely to change the | Low |

\*In some cases, other evidence, such as large all-or-none case series (e.g., jumping from air planes or tall structures), can represent high- or moderate-quality evidence. In such cases, the rationale for the evidence rating exception should be explained by the Work Group and clearly justified.

†"Well-designed, well-executed" refers to studies that directly address the question; use adequate randomization, blinding, and allocation concealment; are adequately powered; use intention-to-treat analyses; and have high follow-up rates

‡Limitations include concerns with the design and execution of a study that result in decreased confidence in the true estimate of the effect. Examples of such limitations include but are not limited to: inadequate randomization, lack of blinding of study participants or outcome assessors, inadequate power, outcomes of interest that are not prespecified for the primary outcomes, low follow-up rates, and findings based on subgroup analyses. Whether the limitations are considered minor or major is based on the number and severity of flaws in design or execution. Rules for determining whether the limitations are considered minor or major and how they will affect rating of the individual studies will be developed collaboratively with the meth-

§Nonrandomized controlled studies refer to intervention studies where assignment to intervention and comparison groups is not random (e.g., quasi-experimental study design).

||Observational studies include prospective and retrospective cohort, case-control, and cross-

NHLBI indicates National Heart, Lung, and Blood Institute; and RCT, randomized controlled

cholesterol (LDL-C) levels with greater ASCVD risk. These studies provided the rationale for RCTs, which in turn demonstrated that lowering cholesterol levels reduced ASCVD events and thereby established a central, causal role of atherogenic cholesterol-containing lipoprotein particles, particularly LDL, in the genesis of CHD and ASCVD.

Other strategies for using drug therapy to reduce ASCVD events have been advocated, including treatto-cholesterol target, lowest-is-best, and risk-based treatment approaches. However, only 1 approach has been evaluated in multiple RCTs—the use of fixed doses of cholesterol-lowering drugs to reduce ASCVD risk. Because the overwhelming body of evidence came from statin

<sup>\*</sup>In most cases, the strength of the recommendation should be closely aligned with the quality of the evidence; however, under some circumstances, there may be valid reasons for making recommendations that are not closely aligned with the quality of the evidence (e.g., strong recommendation when the evidence quality is moderate, such as smoking cessation to reduce cardiovascular disease risk or ordering an ECG as part of the initial diagnostic work-up for a patient presenting with possible MI). Those situations should be limited and the rationale explained clearly by the Work Group.

#### Table 2. What's New in the Guideline?\*

2894

#### 1 Focus on ASCVD Risk Reduction: 4 Statin Benefit Groups

- This guideline is based on a comprehensive set of data from RCTs from which 4 statin benefit groups were identified that focus efforts to reduce ASCVD events in secondary and primary prevention.
- 2. This guideline identifies high-intensity and moderate-intensity statin therapy for use in secondary and primary prevention.
- A New Perspective on LDL-C and/or Non-HDL-C Treatment Goals
   The Expert Panel was unable to find RCT evidence to support
  - continued use of specific LDL-C or non-HDL-C treatment targets.
  - The appropriate intensity of statin therapy should be used to reduce ASCVD risk in those most likely to benefit.
  - Nonstatin therapies, as compared with statin therapy, do not provide acceptable ASCVD risk-reduction benefits relative to their potential for adverse effects in the routine prevention of ASCVD.

#### 3 Global Risk Assessment for Primary Prevention

- This guideline recommends use of the new Pooled Cohort Equations to estimate 10-year ASCVD risk in both white and black men and women.
- By more accurately identifying higher-risk individuals for statin therapy, the guideline focuses statin therapy on those most likely to benefit.
- It also indicates, on the basis of RCT data, those high-risk groups that might not benefit.
- This guideline recommends a discussion between clinicians and patients before initiation of statin therapy.

#### 4 Safety Recommendations

- This guideline used RCTs to identify important safety considerations in individuals receiving treatment of blood cholesterol to reduce ASCVD risk.
- Using RCTs to determine statin adverse effects facilitates understanding of the net benefit from statin therapy.
- This guideline provides expert guidance on management of statin-associated adverse effects, including muscle symptoms.

#### 5 Role of Biomarkers and Noninvasive Tests

 Treatment decisions in selected individuals who are not included in the 4 statin benefit groups may be informed by other factors as recommended by the Risk Assessment Work Group and Blood Cholesterol Expert Panel.

#### 6 Future Updates to the Blood Cholesterol Guideline

- This is a comprehensive guideline for the evidence-based treatment of blood cholesterol to reduce ASCVD risk.
- Future updates will build on this foundation to provide expert guidance on the management of complex lipid disorders and incorporate refinements in risk stratification based on critical review of emerging data.
- RCTs comparing alternative treatment strategies are needed in order to inform future evidence-based guidelines for the optimum ASCVD risk-reduction approach.

\*See Appendix 5, for an expanded discussion of what's new in the guideline.

ASCVD indicates atherosclerotic cardiovascular disease; HDL-C, high-density lipoprotein cholesterol; LDL-C, low-density lipoprotein cholesterol; and RCT, randomized controlled trial.

RCTs, the Expert Panel appropriately focused on these statin RCTs to develop evidence-based guidelines for the reduction of ASCVD risk. We recognize that this represents a significant departure from current strategies. This should not come as a surprise to clinicians. The recent guideline on heart failure has changed long-standing paradigms on the basis of the evidence, and this guideline does as well (5). Future RCTs will be needed to determine the optimal treatment strategy to provide the greatest reduction in ASCVD events with best margin of safety.

The Expert Panel acknowledges that our process did not provide for a comprehensive approach to the detection, evaluation, and treatment of lipid disorders as was done in the prior Adult Treatment Panel III Report (6). However, the present guideline was never intended to be a comprehensive approach to lipid management for purposes other than ASCVD risk reduction. A limited number of expert opinion recommendations were made only when RCT evidence was not present and after a thorough consideration of what the Expert Panel had learned from the RCTs. For the many questions about complex lipid disorders that are beyond the scope of our systematic evidence review, or for which little or no RCT data are available, it is anticipated that clinicians with lipid expertise can contribute to their management.

#### 1.4. Methodology and Evidence Review

Although the Expert Panel was convened before the Institute of Medicine reports on practice guidelines, our evidence-based process followed most of the standards from the Institute of Medicine report, "Clinical Practice Guidelines We Can Trust" (1). The systematic review was limited to RCTs with ASCVD outcomes and systematic reviews and meta-analyses of RCTs with ASCVD outcomes. Observational studies and those with <18 months (CQ1 and CQ2) or <12 months (CQ3) of follow-up were excluded. Support was provided by a methodology contractor and a systematic review and general support contractor and included the following steps:

- The Expert Panel constructed CQs relevant to clinical practice.
- The Expert Panel identified (a priori) inclusion/ exclusion criteria for each CQ.
- An independent contractor developed a literature search strategy, based on inclusion/exclusion criteria, for each CQ.
- An independent contractor executed a systematic electronic search of the published literature from relevant bibliographic databases for each CQ. The date range for the overall literature search was January 1, 1995, through December 1, 2009. However, RCTs with hard ASCVD outcomes of myocardial infarction (MI), stroke, and cardiovascular death published after that date range were eligible for consideration until the Expert Panel began deliberations on relevant recommendations.
- RCTs that met the inclusion criteria and were independently graded as fair or good quality were included in the evidence tables for the consideration of the Expert Panel. RCTs that were graded as poor quality were excluded.
- With the assistance of independent methodologists, this evidence base was used to develop a series of evidence statements graded on the level of the evidence (high, medium, or low).
- The Expert Panel then synthesized the evidence statements into treatment recommendations/summaries

graded as A (strong), B (moderate), C (weak), D (recommend against), E (expert), and N (no recommendation).

- The final evidence statements and treatment recommendations were approved by at least a majority of voting members of the Expert Panel.
- Guideline implementability appraisals, planned and coordinated by the NHLBI Implementation Work Group, were performed to identify and address barriers to guideline implementation.

In addition, the Expert Panel was able to include major RCTs and meta-analyses of RCTs published through July 2013 in our discussion and as part of the process of determining ACC/AHA grading of the NHLBI expert-level recommendations.

#### 2. Overview of the Guideline

The RCTs identified in the systematic evidence review indicated a consistent reduction in ASCVD events from 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitor (statin) therapy in secondary- and primary-prevention populations, with the exception of no ASCVD event reduction when statin therapy was initiated in those with New York Heart Association class II to IV heart failure or those receiving maintenance hemodialysis. The RCTs either compared fixed doses of statins with placebo or untreated controls, or compared fixed doses of higher-intensity statins with moderate-intensity statins. These trials were not designed to evaluate the effect of titrated (dose-adjusted) statin treatment to achieve prespecified LDL-C or non-HDL-C goals.

Therefore, the Expert Panel was unable to find RCT evidence to support titrating cholesterol-lowering drug therapy to achieve target LDL-C or non-HDL-C levels, as recommended by Adult Treatment Panel III (6-8). Notably, the Expert Panel did find RCT evidence that use of therapy (e.g., niacin) to additionally lower non-HDL-C, once an LDL-C target was achieved, did not further reduce ASCVD outcomes (9). The Expert Panel also found extensive RCT evidence that the appropriate intensity of statin therapy should be used to reduce ASCVD risk in those most likely to benefit. The work of the Expert Panel was informed by the reports of the Lifestyle Management (10) and Risk Assessment Work Groups (11) (Figure 1). A summary of the major recommendations for the treatment of cholesterol to reduce ASCVD risk is provided in Table 3.

### 2.1. Lifestyle as the Foundation for ASCVD Risk-Reduction Efforts

It must be emphasized that lifestyle modification (i.e., adhering to a heart-healthy diet, regular exercise habits, avoidance of tobacco products, and maintenance of a healthy weight) remains a crucial component of health promotion and ASCVD risk reduction, both prior to and in concert with the use of cholesterol-lowering drug therapies. Healthy diet or lifestyle modifications were recommended as background therapy for the RCTs of cholesterol-lowering drug therapy. See the "2013 AHA/ACC Guideline on Lifestyle Management to Reduce Cardiovascular Risk" (10) for lifestyle recommendations for healthy adults. Drug therapy for lifestyle-related risk factors such as hypertension is often needed and smoking should be avoided.



Figure 1. Overview of the Expert Panel's Guideline

2896

### Table 3. Summary of Key Recommendations for the Treatment of Blood Cholesterol to Reduce ASCVD Risk in Adults (See Tables 4, 8, 9, and 10 for the complete recommendations; and Table 5 for definition of statin intensity)

| Recommendations | ACC/AHA COR | ACC/AHA LOE |
|---|---|---|
| A. Heart-healthy lifestyle habits should be encouraged for all individuals | | |
| B. The appropriate intensity of statin therapy should be initiated or continued: | | |
| 1. Clinical ASCVD* | | |
| a. Age $\leq 75$ y and no safety concerns: High-intensity statin | 1 | Α |
| b. Age >75 y or safety concerns: Moderate-intensity statin | | A |
| 2. Primary prevention – Primary LDL-C ≥190 mg/dL | | |
| a. Rule out secondary causes of hyperlipidemia (Table 6) | 1 | В |
| b. Age ≥21 y: High-intensity statin | 1 | В |
| c. Achieve at least a 50% reduction in LDL-C | lla | В |
| d. LDL-C lowering nonstatin therapy may be considered to further reduce LDL-C | IIb | С |
| 3. Primary prevention—Diabetes 40–75 years of age and LDL-C 70–189 mg/dL | | |
| a. Moderate-intensity statin | 1 | Α |
| b. Consider high-intensity statin when $\geq$ 7.5% 10-y ASCVD risk using the Pooled Cohort Equations $\dagger$ | lla | В |
| 4. Primary prevention – No diabetes 40–75 years of age and LDL-C 70–189 mg/dL | | |
| a. Estimate 10-y ASCVD risk using the Risk Calculator based on the Pooled Cohort Equations† in those NOT receiving a statin; | 1 | В |
| estimate risk every 4-6 y | | |
| b. To determine whether to initiate a statin, engage in a clinician-patient discussion of the potential for ASCVD risk reduction, | lla | С |
| adverse effects, drug-drug interactions, and patient preferences | | |
| <ul> <li>c. Re-emphasize heart-healthy lifestyle habits and address other risk factors</li> <li>i. ≥7.5% 10-y ASCVD risk: Moderate- or high-intensity statin</li> </ul> | 1 | Α |
| ii. 5 to <7.5% 10-y ASCVD risk: Consider moderate-intensity statin | lla | B |
| iii. Other factors may be considered‡: LDL-C ≥160 mg/dL, family history of premature ASCVD, hs-CRP ≥2.0 mg/L, | IIb | C |
| CAC score $\geq$ 300 Agaston units, ABI <0.9, or lifetime ASCVD risk | 110 | · |
| 5. Primary prevention when LDL-C <190 mg/dL and age <40 or >75 y, or <5% 10-y ASCVD risk | IIb | С |
| a. Statin therapy may be considered in selected individuals‡ | | |
| 6. Statin therapy is not routinely recommended for individuals with NYHA class II-IV heart failure or who are receiving | | |
| maintenance hemodialysis | | |
| C. Regularly monitor adherence to lifestyle and drug therapy with lipid and safety assessments | | |
| 1. Assess adherence, response to therapy, and adverse effects within 4-12 wk following statin initiation or change in therapy | 1 | Α |
| a. Measure a fasting lipid panel | ı | Α |
| b. Do not routinely monitor ALT or CK unless symptomatic | lla | С |
| c. Screen and treat type 2 diabetes according to current practice guidelines. Heart-healthy lifestyle habits should be encouraged | 1 | В |
| to prevent progression to diabetes | | - |
| d. Anticipated therapeutic response: approximately ≥50% reduction in LDL-C from baseline for high-intensity statin and<br>30% to <50% for moderate-intensity statin | lla | В |
| i. Insufficient evidence for LDL-C or non-HDL-C treatment targets from RCTs | | |
| ii. For those with unknown baseline LDL-C, an LDL-C <100 mg/dL was observed in RCTs of high-intensity statin therapy | | |
| e. Less than anticipated therapeutic response: i. Reinforce improved adherence to lifestyle and drug therapy | | Α |
| ii. Evaluate for secondary causes of hyperlipidemia if indicated (Table 6) | | Δ |
| iii. Increase statin intensity, or if on maximally-tolerated statin intensity, consider addition of nonstatin therapy in selected | IIb | C |
| high-risk individuals§ | 110 | C |
| f. Regularly monitor adherence to lifestyle and drug therapy every 3–12 mo once adherence has been established. Continue | 1 | A |
| assessment of adherence for optimal ASCVD risk reduction and safety | | |
| assessment of authorities for optimal ASCVD fish reduction and safety | 1 | В |
| D. In individuals intolerant of the recommended intensity of statin therapy, use the maximally tolerated intensity of | | |
| <ol><li>In individuals intolerant of the recommended intensity of statin therapy, use the maximally tolerated intensity of<br/>statin.</li></ol> | | |
| D. In individuals intolerant of the recommended intensity of statin therapy, use the maximally tolerated intensity of | lla | В |

\*Clinical ASCVD includes acute coronary syndromes, history of MI, stable or unstable angina, coronary or other arterial revascularization, stroke, TIA, or peripheral arterial disease presumed to be of atherosclerotic origin.

†Estimated 10-year or "hard" ASCVD risk includes first occurrence of nonfatal MI, CHD death, and nonfatal and fatal stroke as used by the Risk Assessment Work Group in developing the Pooled Cohort Equations (http://my.americanheart.org/cvriskcalculator and http://www.cardiosource.org/en/Science-And-Quality/Practice-Quidelines-and-Quality-Standards/2013-Prevention-Quideline-Tools.aspx). †These factors may include primary LDL-C ≥160 mg/dL or other evidence of genetic hyperlipidemias; family history of premature ASCVD with onset <55 years of age in a first-degree male relative; hs-CRP ≥2 mg/L; CAC score ≥300 Agastson units or ≥75th percentile for age, sex, and ethnicity (for additional information, see http://www.mesa-nhlbi.org/CACReference.aspx); ABI <0.9; or lifetime risk of ASCVD. Additional factors that might aid in individual risk assessment could be identified in the future.

§High-risk individuals include those with clinical ASCVD, an untreated LDL-C ≥190 mg/dL suggesting genetic hypercholesterolemia, or individuals with diabetes 40 to 75 years of age and LDL-C 70 to 189 mg/dL.

ABI indicates ankle-brachial index; ACC, American College of Cardiology; AHA, American Heart Association; ALT, alanine aminotransferase, a test of hepatic function; ASCVD, atherosclerotic cardiovascular disease; CAC, coronary artery calcium; CHD, coronary heart disease; CK, creatine kinase, a test of muscle injury; COR, Class of Recommendation; HDL-C, high-density lipoprotein cholesterol; hs-CRP, high-sensitivity C-reactive protein; LDL-C, low-density lipoprotein cholesterol; LOE, Level of Evidence; NHLBI, National Heart, Lung, and Blood Institute; NYHA, New York Heart Association; RCTs, randomized controlled trials; and TIA, transient ischemic attack.

#### 2.2. Initiation of Statin Therapy

The Expert Panel found extensive and consistent evidence supporting the use of statins for the prevention of ASCVD in many higher-risk primary- and all secondary-prevention individuals without New York Heart Association class II-IV heart failure who were not receiving hemodialysis. In the RCTs reviewed, initiation of moderate-intensity therapy (lowering LDL-C by approximately 30% to <50%) or high-intensity statin therapy (lowering LDL-C by approximately  $\geq 50\%$ ) is a critical factor in reducing ASCVD events. Moreover, statin therapy reduces ASCVD events across the spectrum of baseline LDL-C levels ≥70 mg/dL. In addition, the relative reduction in ASCVD risk is consistent for primary and secondary prevention and for various patient subgroups. Of note, the absolute reduction in ASCVD events is proportional to baseline absolute ASCVD risk. Therefore, statin therapy is recommended for individuals at increased ASCVD risk who are most likely to experience a net benefit in terms of the potential for ASCVD risk reduction and the potential for adverse effects (Table 3;

On the basis of this large and consistent body of evidence, 4 major statin benefit groups were identified for whom the ASCVD risk reduction clearly outweighs the risk of adverse events based on a strong body of evidence. These are 1) secondary prevention in individuals with clinical ASCVD, 2) primary prevention in individuals with primary elevations of LDL-C ≥190 mg/dL, 3) primary prevention in individuals with diabetes 40 to 75 years of age who have LDL-C 70 to 189 mg/dL, and 4) primary prevention in individuals without diabetes and with estimated 10-year ASCVD risk ≥7.5%, 40 to 75 years of age who have LDL-C 70 to 189 mg/dL. Moderate evidence supports the use of statins for primary prevention in individuals with 5% to <7.5% 10-year ASCVD risk, 40 to 75 years of age with LDL-C 70 to 189 mg/dL. Selected individuals with <5% 10-year ASCVD risk, or <40 or >75 years of age may also benefit from statin therapy. Clinicians and patients should engage in a discussion of the potential for ASCVD risk-reduction benefits, adverse effects, drug-drug interactions, and consider patient preferences for treatment. This discussion also provides the opportunity to re-emphasize healthy-lifestyle habits and address other risk factors.

Clinical ASCVD is defined by the inclusion criteria for the secondary-prevention statin RCTs (acute coronary syndromes, a history of MI, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack, or peripheral arterial disease presumed to be of atherosclerotic origin). For primary prevention in individuals without clinical ASCVD or diabetes who have an LDL-C 70 to 189 mg/dL, the estimated absolute 10-year risk of ASCVD (defined as nonfatal MI, CHD death, or nonfatal and fatal stroke)

should be used to guide the initiation of statin therapy. The 10-year ASCVD risk should be estimated with the Pooled Cohort Equations (Section 4.7). For the primary prevention of ASCVD in individuals with diabetes (diabetes mellitus type 1 and type 2), estimated 10-year ASCVD risk can also be used to guide the intensity of statin therapy. For those with clinical ASCVD or with LDL-C ≥190 mg/dL who are already in a statin benefit group, it is not appropriate to estimate 10-year ASCVD risk. In primary prevention, additional factors may influence ASCVD risk in those for whom a risk-based decision is unclear. These include a primary LDL-C ≥160 mg/dL or other evidence of genetic hyperlipidemias, family history of premature ASCVD with onset <55 years of age in a first-degree male relative or <65 years of age in a first-degree female relative, highsensitivity C-reactive protein ≥2 mg/L, coronary artery calcium score  $\geq$ 300 Agatston units or  $\geq$ 75th percentile for age, sex, and ethnicity (for additional information, see http://www.mesa-nhlbi.org/CACReference.aspx.), anklebrachial index <0.9, and elevated lifetime risk of ASCVD.

The findings support the use of statins to prevent both nonfatal and fatal ASCVD events. Such an approach can reduce the large burden of disability from nonfatal stroke (for which women are at higher risk than men) and nonfatal CHD events. Primary and secondary prevention of ASCVD with statins can positively impact rising healthcare costs. In addition, a high level of evidence was found that statins reduce total mortality in individuals with a history of prior ASCVD events (e.g., secondaryprevention settings). In individuals with no prior history of ASCVD events (e.g., primary-prevention settings), there is moderate evidence that statins reduce total mortality in individuals at increased ASCVD risk. It should be noted that 2 meta-analyses published after the completion of the Expert Panel's systematic review provide strong evidence that statins reduce total mortality in primary prevention (12,13).

#### 3. Critical Questions and Conclusions

#### 3.1. Identification of CQs

Although limited to 3 CQs, these questions were considered the most important to answer in order to identify whom to treat and with what treatment(s) and to consider how intensively the treatments should be used. The first 2 CQs evaluated the evidence for LDL-C and non-HDL-C goals for the secondary and primary prevention of ASCVD with cholesterol-lowering drug therapy. Titration to specific LDL-C goals has been considered a fundamental therapeutic strategy in deciding on the adequacy of cholesterol-lowering therapy for secondary and primary prevention. Therefore, a comprehensive systematic review



Figure 2. Summary of Statin Initiation Recommendations for the Treatment of Blood Cholesterol to Reduce ASCVD Risk in Adults (See Figures 3, 4, and 5 for More Detailed Management Information)

Colors correspond to the Classes of Recommendation in Table 1. Assessment of the potential for benefit and risk from statin therapy for ASCVD prevention provides the framework for clinical decision making incorporating patient preferences.

†The Pooled Cohort Equations can be used to estimate 10-year ASCVD risk in individuals with and without diabetes. The estimator within this application should be used to inform decision making in primary prevention patients not on a statin.

‡Consider moderate-intensity statin as more appropriate in low-risk individuals.

 $\S$ For those in whom a risk assessment is uncertain, consider factors such as primary LDL-C  $\ge$ 160 mg/dL or other evidence of genetic hyperlipidemias, family history of premature ASCVD with onset <55 years of age in a first-degree male relative or <65 years of age in a first-degree female relative, hs-CRP  $\ge$ 2 mg/L, CAC score  $\ge$ 300 Agatston units, or  $\ge$ 75th percentile for age, sex, and ethnicity (for additional information, see http://www.mesa-nhlbi.org/CACReference.aspx), ABI <0.9, or lifetime risk of ASCVD. Additional factors that may aid in individual risk assessment may be identified in the future.

 $\parallel$ Potential ASCVD risk-reduction benefits. The absolute reduction in ASCVD events from moderate- or high-intensity statin therapy can be approximated by multiplying the estimated 10-year ASCVD risk by the anticipated relative-risk reduction from the intensity of statin initiated ( $\sim$  30% for moderate-intensity statin or  $\sim$  45% for high-intensity statin therapy). The net ASCVD risk-reduction benefit is estimated from the number of potential ASCVD events prevented with a statin, compared to the number of potential excess adverse effects. Petential adverse effects. The excess risk of diabetes is the main consideration in  $\sim$  0.1 excess cases per 100 individuals treated with a moderate-intensity statin for 1 year and  $\sim$  0.3 excess cases per 100 individuals treated with a high-intensity statin for 1 year. In RCTs, both statin-treated and placebo-treated participants experienced the same rate of muscle symptoms. The actual rate of statin-related muscle symptoms in the clinical population is unclear. Muscle symptoms attributed to statin therapy should be evaluated (see Table 8. Safety Recommendation 8).

ABI indicates ankle-brachial index; ASCVD, atherosclerotic cardiovascular disease; CAC, coronary artery calcium; hs-CRP, high-sensitivity C-reactive protein; LDL-C, low-density lipoprotein cholesterol; MI, myocardial infarction; and RCT, randomized controlled trial.

<sup>\*</sup>Percent reduction in LDL-C can be used as an indication of response and adherence to therapy, but is not in itself a treatment goal.

of the evidence base supporting this concept was essential. The third CQ had several objectives:

- Identify groups of patients who will benefit from pharmacological treatment,
- Define the pharmacological treatment(s) for which there is the best evidence of net benefit, and
- Provide guidance on the appropriate intensity of pharmacological treatment to reduce ASCVD risk.

### 3.1.1. CQ1: LDL-C and Non-HDL-C Goals in Secondary Prevention

### CQ1: What is the evidence for LDL-C and non-HDL-C goals for the secondary prevention of ASCVD?

The Expert Panel reviewed 19 RCTs to answer CQ1. Although CQ1 is supported conceptually by an extrapolation of observational studies and observational data from RCTs, no data were identified for treatment or titration to a specific LDL-C goal in adults with clinical ASCVD. The majority of studies confirming the efficacy of cholesterol reduction in improving clinical outcomes in patients with clinical ASCVD used a single fixed-dose statin to lower LDL-C levels. In the 4S trial, 37% had the dose of simvastatin raised from 20 mg/d to 40 mg/d to achieve a total cholesterol level <200 mg/dL (16). The Expert Panel was unable to find any RCTs that evaluated titration of all individuals in a treatment group to specific LDL-C targets <100 mg/dL or <70 mg/dL, nor were any RCTs comparing 2 LDL-C treatment targets identified. No statin RCTs reporting on-treatment non-HDL-C levels were identified. (In CQ3, statin-nonstatin combination therapy was evaluated.)

### 3.1.2. CQ2: LDL-C and Non-HDL-C Goals in Primary Prevention

### CQ2: What is the evidence for LDL-C and non-HDL-C goals for the primary prevention of ASCVD?

The Expert Panel reviewed 6 RCTs. The 4 studies confirming the efficacy of cholesterol reduction in improving clinical outcomes in patients without ASCVD used fixeddose statin therapy to lower LDL-C levels. In the AFCAPS-TEXCAPS (Air Force/Texas Coronary Atherosclerosis Prevention Study) trial (17), in 50% of participants, the lovastatin dose was raised from 20 mg to 40 mg to achieve an LDL-C level <110 mg/dL. In the MEGA (Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese) trial (18), the dose of pravastatin could be uptitrated from 10 mg to 20 mg to achieve a total cholesterol level <220 mg/dL. The Expert Panel did not find any RCTs that evaluated titration of all individuals in a treatment group to specific LDL-C targets <100 mg/dL or <70 mg/dL, nor were any RCTs comparing 2 LDL-C treatment targets identified. No trials reported on-treatment non-HDL-C levels.

### 3.1.3. CQ3: Efficacy and Safety of Cholesterol-Lowering Medications

#### CQ3: For primary and secondary prevention, what is the impact on lipid levels, effectiveness, and safety of specific cholesterol-modifying drugs used for lipid management in general and in selected subgroups?

The populations examined included primary-prevention adult patients who could not have a diagnosis of CHD or cardiovascular disease. Interventions included pharmacotherapy with single-drug therapies or combination-drug therapies with any drug therapy used for treating blood cholesterol, including statins, fibrates (fenofibrate, gemfibrozil), nicotinic acid (niacin in immediate-, slow-, or extended-release form), bile acid sequestrants, ezetimibe, omega-3 fatty acids (also called marine fatty acids, including eicosapentaenoic acid alone, docosahexanoic acid alone, eicosapentaenoic acid plus docosahexanoic acid, and alpha-linolenic acid). There were no ASCVD outcomes identified for plant sterols, sterol esters, stanols, or stanol esters. A single ASCVD outcomes trial (19) used Xuezhikang, an extract from red yeast Chinese rice, which was not available in the United States during the timeframe for evidence review, so no recommendations were made regarding its use.

The recommendations synthesize the evidence retrieved for answering CQ3, along with the evidence from the trials included in CQ1 and CQ2, to guide the use of cholesterol-lowering drugs for secondary or primary prevention of ASCVD.

#### 4. Statin Treatment: Recommendations

For each recommendation, the grades of the recommendation by both the NHLBI and ACC/AHA methods are provided. Major treatment recommendations are listed in Table 4, and statin intensities are defined in Table 5. The safety (statin and nonstatin) recommendations are in Section 5. A complete listing of the evidence statements supporting each recommendation, along with the references, is provided in Appendix 4.

### **4.1. Intensity of Statin Therapy in Primary and Secondary Prevention**

The Expert Panel defines the intensity of statin therapy on the basis of the average expected LDL-C response to a specific statin and dose. "High-intensity," "moderate-intensity," and "low-intensity" statin therapy definitions were derived from the systematic reviews for CQ1 and CQ2. The basis for differentiation among specific statins and doses arose from the RCTs included in CQ1, where there was a high level of evidence that high-intensity statin therapy with atorvastatin 40 mg to 80 mg reduced ASCVD risk more than moderate-intensity

Table 4. Recommendations for Treatment of Blood Cholesterol to Reduce Atherosclerotic Cardiovascular Risk in Adults—Statin Treatment (High, Moderate, and Low Statin Intensities are Defined in Table 5)

| Recommendations | NHLBI Grade | NHLBI Evidence<br>Statements | ACC/AHA COR | ACC/AHA LOE |
|---|---|---|---|---|
| Treatment Targets | | | , | |
| <ol> <li>The Expert Panel makes no recommendations for or<br/>against specific LDL-C or non-HDL-C targets for the<br/>primary or secondary prevention of ASCVD.</li> </ol> | N (No recommendation) | 1-4 | _ | _ |
| Secondary Prevention | | | | |
| L. High-intensity statin therapy should be initiated or<br>continued as first-line therapy in women and men<br>≤75 years of age who have clinical ASCVD*, unless<br>contraindicated. | A (Strong) | 1,6-8,10-23,26-28 | ı | A |
| 2. In individuals with clinical ASCVD* in whom high-intensity statin therapy would otherwise be used, when high-intensity statin therapy is contraindicated† or when characteristics predisposing to statin-associated adverse effects are present, moderate-intensity statin should be used as the second option if tolerated (Table 8 for Safety of Statins, Recommendation 1). | A (Strong) | 13-22,24,27,28 | 1 | А |
| 3. In individuals with clinical ASCVD >75 years of age, it is reasonable to evaluate the potential for ASCVD risk-reduction benefits and for adverse effects and drug-drug interactions and to consider patient preferences when initiating a moderate- or high-intensity statin. It is reasonable to continue statin therapy in those who are tolerating it. Primary Prevention in Individuals ≥21 Years of Age With LD | E (Expert Opinion) | _ | lla | <b>B</b><br>(16,20-43) |
| _ | B (Moderate) | 75 | I‡ | В |
| L. Individuals with LDL-C ≥190 mg/dL or triglycerides<br>≥500 mg/dL should be evaluated for secondary causes<br>of hyperlipidemia (Table 6). | b (Woderate) | 13 | •+ | (44,45) |
| <ol> <li>Adults ≥21 years of age with primary LDL-C ≥190 mg/dL should be treated with statin therapy (10-year ASCVD risk estimation is not required):</li> <li>Use high-intensity statin therapy unless contraindicated.</li> <li>For individuals unable to tolerate high-intensity statin therapy, use the maximum tolerated statin intensity.</li> </ol> | B (Moderate) | 6,19,28,33-35,37,38 | I§ | В |
| <ol> <li>For individuals ≥21 years of age with an untreated<br/>primary LDL-C ≥190 mg/dL, it is reasonable to intensify<br/>statin therapy to achieve at least a 50% LDL-C reduction.</li> </ol> | E (Expert Opinion) | _ | lla | <b>B</b><br>(20,46-50) |
| 4. For individuals ≥21 years of age with an untreated primary LDL-C ≥190 mg/dL, after the maximum intensity of statin therapy has been achieved, addition of a non-statin drug may be considered to further lower LDL-C. Evaluate the potential for ASCVD risk-reduction benefits, adverse effects, and drug-drug interactions, and consider patient preferences. | E (Expert Opinion) | _ | IIb | <b>C</b> (51) |
| Primary Prevention in Individuals With Diabetes and LDL-C | | | | |
| <ol> <li>Moderate-intensity statin therapy should be initiated<br/>or continued for adults 40–75 years of age with diabetes.</li> </ol> | A (Strong) | 19,29-34,40 | 1 | Α |
| <ol> <li>High-intensity statin therapy is reasonable for adults<br/>40–75 years of age with diabetes with a ≥7.5%<br/>estimated 10-year ASCVD risk unless contraindicated.</li> </ol> | E (Expert Opinion) | _ | lla | <b>B</b><br>(49,52) |
| 3. In adults with diabetes, who are <40 years of age or<br>>75 years of age, or with LDL <70 mg/dL it is reasonable to evaluate the potential for ASCVD benefits and for adverse effects and drug-drug interactions and to consider patient preferences when deciding to initiate, continue, or intensify statin therapy. | E (Expert Opinion) | _ | lla | <b>C</b><br>(53-62) |

Continued on the next page

**Table 4. Continued** 

| | | NHLBI Evidence | | |
|---|---|---|---|---|
| Recommendations | NHLBI Grade | Statements | ACC/AHA COR | ACC/AHA LOE |
| Primary Prevention in Individuals Without Diabetes and Wit | <b>.</b> , | | | _ |
| <ol> <li>The Pooled Cohort Equations should be used to estimate<br/>10-year ASCVD risk for individuals with LDL-C 70-189<br/>mg/dL without clinical ASCVD* to guide initiation of<br/>statin therapy for the primary prevention of ASCVD.</li> </ol> | E (Expert Opinion) | _ | • | <b>B</b><br>(11) |
| <ol> <li>Adults 40-75 years of age with LDL-C 70-189 mg/dL,<br/>without clinical ASCVD* or diabetes, and with an<br/>estimated 10-year ASCVD∥ risk ≥7.5% should be treated<br/>with moderate- to high-intensity statin therapy.</li> </ol> | A (Strong) | 28,34-36,38,42-44,<br>47,49-56,76 | ı | А |
| <ol> <li>It is reasonable to offer treatment with a moderate-<br/>intensity statin to adults 40–75 years of age, with LDL-C<br/>70–189 mg/dL, without clinical ASCVD* or diabetes, and<br/>with an estimated 10-year ASCVD∥ risk of 5% to &lt;7.5%.</li> </ol> | C (Weak) | 28,34-36,38,42-44,<br>47,49-56,76 | lla | В |
| 4. Before initiation of statin therapy for the primary prevention of ASCVD in adults with LDL-C 70–189 mg/dL without clinical ASCVD* or diabetes, it is reasonable for clinicians and patients to engage in a discussion that considers the potential for ASCVD risk-reduction benefits and for adverse effects and drug-drug interactions, as well as patient preferences for treatment. | E (Expert Opinion) | _ | lla | <b>C</b><br>(63) |
| 5. In adults with LDL-C <190 mg/dL who are not otherwise identified in a statin benefit group, or for whom after quantitative risk assessment a risk-based treatment decision is uncertain, additional factors¶ may be considered to inform treatment decision making. In these individuals, statin therapy for primary prevention may be considered after evaluation of the potential for ASCVD risk-reduction benefits, adverse effects, and drugdrug interactions and consider patient preferences. | E (Expert Opinion) | _ | IIb | <b>c</b><br>(11,13) |
| Heart Failure and Hemodialysis | | | | |
| 1. The Expert Panel makes no recommendations regarding the initiation or discontinuation of statins in patients with NYHA class II-IV ischemic systolic heart failure or in patients on maintenance hemodialysis. | N (No Recommendation) | 71,72 | _ | _ |

\*Clinical ASCVD includes acute coronary syndromes, history of MI, stable or unstable angina, coronary or other arterial revascularization, stroke, TIA, or peripheral arterial disease presumed to be of atherosclerotic origin.

†Contraindications, warnings, and precautions are defined for each statin according to the manufacturer's prescribing information (64–70).

‡Individuals with secondary causes of hyperlipidemia were excluded from RCTs reviewed. A triglyceride level ≥500 mg/dL was an exclusion criterion for almost all RCTs. Therefore, ruling out secondary causes is necessary to avoid inappropriate statin therapy.

§No RCTs included only individuals with LDL-C  $\geq$ 190 mg/dL. However, many trials did include individuals with LDL-C  $\geq$ 190 mg/dL, and all of these trials consistently demonstrated a reduction in ASCVD events. In addition, the Cholesterol Treatment Trialists meta-analyses have shown that each 39-mg/dL reduction in LDL-C with statin therapy reduced ASCVD events by 22%, and the relative reductions in ASCVD events were consistent across the range of LDL-C levels. Therefore, individuals with primary LDL-C  $\geq$ 190 mg/dL should be treated with statin therapy.

||Estimated 10-year or "hard" ASCVD risk includes first occurrence of nonfatal MI, coronary heart disease death, and nonfatal and fatal stroke as used by the Risk Assessment Work Group in developing the Pooled Cohort Equations.

¶These factors may include primary LDL-C  $\geq$ 160 mg/dL or other evidence of genetic hyperlipidemias; family history of premature ASCVD with onset <55 years of age in a first-degree male relative or <65 years of age in a first-degree female relative; high-sensitivity C-reactive protein  $\geq$ 2 mg/L; CAC score  $\geq$ 300 Agatston units or  $\geq$ 75th percentile for age, sex, and ethnicity (for additional information, see http://www.mesa-nhlbi.org/CACReference.aspx); ABI <0.9; or lifetime risk of ASCVD. Additional factors that might aid in individual risk assessment could be identified in the future.

ABI indicates ankle-brachial index; ACC, American College of Cardiology; AHA, American Heart Association; ASCVD, atherosclerotic cardiovascular disease; CAC, coronary artery calcium; COR, Class of Recommendation; HDL-C, high-density lipoprotein cholesterol; LDL-C, low-density lipoprotein cholesterol; LOE, Level of Evidence; NHLBI, National Heart, Lung, and Blood Institute; NYHA, New York Heart Association; RCTs, randomized controlled trials; TIA, transient ischemic attack; and —, not applicable.

statin therapy with atorvastatin 10 mg, pravastatin 40 mg, or simvastatin 20 mg to 40 mg twice daily. Classifying specific statins and doses by the percent reduction in LDL-C level is based on evidence that the relative reduction in ASCVD risk from statin therapy is related to the degree by which LDL-C is lowered. However, no variation in the relative reduction in ASCVD risk was observed after the data were adjusted for LDL-C reduction. Furthermore, there is no differentiation between the specific statins and doses used in primary- and secondary-prevention RCTs, according to a high level of evidence that statins reduce ASCVD risk similarly in both populations.

Percent reductions in LDL-C for a specific statin and dose were calculated for the RCTs included in individual meta-analyses conducted by the Cholesterol Treatment Trialists (CTT) in 2010 (20), in which statin therapy reduced ASCVD events. High-intensity statin therapy on average lowers LDL-C by approximately ≥50%, moderate-intensity statin therapy lowers LDL-C by approximately 30% to <50%, and lower-intensity statin therapy lowers LDL-C by <30% (Table 5).

#### 4.2. LDL-C and Non-HDL-C Treatment Goals

The Expert Panel did not find evidence to support titrating cholesterol-lowering drug therapy to achieve optimal

Table 5. High-, Moderate-, and Low-Intensity Statin Therapy (Used in the RCTs Reviewed by the Expert Panel)\*

| High-Intensity Statin Therapy | Moderate-Intensity Statin Therapy | Low-Intensity Statin Therapy |
|---|---|---|
| Daily dose lowers LDL-C, on average, | Daily dose lowers LDL-C, on average, | Daily dose lowers LDL-C, |
| by approximately ≥50% | by approximately 30% to $<$ 50% | on average, by $<$ 30% |
| Atorvastatin (40†)–80 mg | Atorvastatin 10 (20) mg | Simvastatin 10 mg |
| Rosuvastatin 20 (40) mg | Rosuvastatin (5) 10 mg | Pravastatin 10–20 mg |
| | Simvastatin 20–40 mg‡ | Lovastatin 20 mg |
| | Pravastatin 40 (80) mg | Fluvastatin 20–40 mg |
| | Lovastatin 40 mg | Pitavastatin 1 mg |
| | Fluvastatin XL 80 mg | |
| | Fluvastatin 40 mg BID | |
| | Pitavastatin 2–4 mg | |

Boldface type indicates specific statins and doses that were evaluated in RCTs (16–18,46–49,64–75,77) included in CQ1, CQ2, and the Cholesterol Treatment Trialists 2010 meta-analysis included in CQ3 (20). All of these RCTs demonstrated a reduction in major cardiovascular events. Italic type indicates statins and doses that have been approved by the FDA but were not tested in the RCTs reviewed.

\*Individual responses to statin therapy varied in the RCTs and should be expected to vary in clinical practice. There might be a biological basis for a less-than-average response.

†Evidence from 1 RCT only: down-titration if unable to tolerate atorvastatin 80 mg in the IDEAL (Incremental Decrease through Aggressive Lipid Lowering) study (47).

‡Although simvastatin 80 mg was evaluated in RCTs, initiation of simvastatin 80 mg or titration to 80 mg is not recommended by the FDA because of the increased risk of myopathy, including

BID indicates twice daily; CQ, critical question; FDA, Food and Drug Administration; LDL-C, low-density lipoprotein cholesterol; and RCTs, randomized controlled trials.

LDL-C or non-HDL-C levels because the clinical trials were essentially fixed-dose trials (CQ1 and CQ2). Dosage increases did occur in a few RCTs with the intent of maximizing statin therapy. Therefore, these were not truly tests of defining optimal goals for LDL-C in primary and secondary prevention because not all individuals in the statin treatment groups received drug therapy titrated to achieve a specific LDL-C or non-HDL-C goal, nor were specific treatment targets compared. One RCT in CQ3 was identified that showed no additional ASCVD event reduction from the addition of nonstatin therapy to further lower non-HDL-C levels once an LDL-C goal had been reached. In AIM-HIGH (Atherothrombosis Intervention in Metabolic Syndrome With Low HDL/ High Triglycerides and Impact on Global Health Outcomes), the additional reduction in non-HDL-C levels (as well as further reductions in apolipoprotein B, lipoprotein[a], and triglycerides in addition to HDL-C increases) with niacin therapy did not further reduce ASCVD risk in individuals treated to LDL-C levels of 40 to 80 mg/dL (9).

Therefore, given the absence of data on titration of drug therapy to specific goals, no recommendations are made for or against specific LDL-C or non-HDL-C goals for the primary or secondary prevention of ASCVD.

#### 4.3. Secondary Prevention

Women and men with clinical ASCVD (defined from the RCT inclusion criteria as acute coronary syndromes; history of MI, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack, or peripheral arterial disease presumed to be of atherosclerotic origin) arterial revascularization, stroke, transient ischemic attack, or peripheral arterial disease presumed to be of atherosclerotic origin are at increased risk for recurrent ASCVD and ASCVD death. An extensive body of evidence demonstrates that high-intensity statin therapy reduces ASCVD events more than moderate-intensity statin therapy (Table 4) in individuals with clinical ASCVD.

High-intensity statin therapy should be initiated for adults ≤75 years of age with clinical ASCVD who are not receiving statin therapy, or the intensity should be increased in those receiving a low- or moderate-intensity statin, unless they have a history of intolerance to high-intensity statin therapy or other characteristics that could influence safety (Section 5). This is consistent with RCT data. In 2 trials, patients were previously treated with a moderately intensive statin (46,47), and in 2 trials, 75% to 97% of patients had not received prior statin therapy (48,78). The high-intensity statins atorvastatin 80 mg and rosuvastatin 20 mg daily reduce LDL-C ≥50% on average and have been shown to reduce ASCVD events in RCTs.

Although atorvastatin 40 mg reduces LDL-C by approximately ≥50%, this dose was used in only 1 RCT if the participant was unable to tolerate atorvastatin 80 mg/dL. Whether an individual receiving atorvastatin 40 mg should be uptitrated to atorvastatin 80 mg should be based on the potential for an ASCVD risk-reduction benefit and the potential for adverse effects, drug-drug interactions, and consider patient preferences.

In individuals with clinical ASCVD in whom highintensity statin therapy would otherwise be used, either when high-intensity statin therapy is contraindicated or when characteristics predisposing to statin-associated adverse effects are present, moderate-intensity statin should be used as the second option, if tolerated (Section 5). In the relatively few individuals >75 years of age who were included in RCTs of high- versus moderate-intensity statin therapy, there was no clear evidence of an additional reduction in ASCVD events from high-intensity statin therapy. In contrast, individuals >75 years of age did experience a reduction in ASCVD events in the trials of mostly moderateintensity statin therapy, as compared with control. Therefore, moderate-intensity statin therapy should be considered for individuals >75 years of age with clinical ASCVD. However, in acknowledgment that older participants in RCTs were likely to be healthier than many older individuals in the general population, the use of statin therapy should be individualized



Figure 3. Initiating Statin Therapy in Individuals With Clinical ASCVD

Colors correspond to the Classes of Recommendation in Table 1.

ALT indicates alanine transaminase; ASCVD, atherosclerotic cardiovascular disease; CK, creatine kinase; FH, familial hypercholesterolemia; LDL-C, low-density lipoprotein cholesterol; and ULN, upper limit of normal.

in persons >75 years of age with *clinical* ASCVD, according to the potential for ASCVD risk-reduction benefits, adverse effects, drug-drug interactions, and consider patient preferences. The Expert Panel considers it reasonable to continue statin therapy in persons >75 years of age who have *clinical* ASCVD and are tolerating statin therapy.

The flow diagram for the initiation and management of statin therapy in individuals with *clinical* ASCVD is provided in Figure 3.

#### 4.4. Primary Prevention in Individuals ≥21 Years of Age With LDL-C ≥190 mg/dL

This guideline recognizes that individuals ≥21 years of age with primary, severe elevations of LDL-C (≥190 mg/dL) have a high lifetime risk for ASCVD events. This is due to their lifetime exposure to markedly elevated LDL-C levels arising from genetic causes. Thus, at age 21, these individuals should receive statin therapy if they have not already been diagnosed and treated before this age. Although in most clinical trials individuals with LDL-C ≥190 mg/dL were not included because of their need for treatment, extensive evidence shows that each 39-mg/dL reduction in LDL-C by statin therapy reduces ASCVD risk by about 20%. Patients with primary elevations of LDL-C ≥190 mg/dL require even more substantial reductions in their LDL-C levels and intensive management

Table 6. Secondary Causes of Hyperlipidemia Most Commonly Encountered in Clinical Practice

| Secondary Cause | Elevated LDL-C | Elevated<br>Triglycerides |
|---|---|---|
| Diet | Saturated or <i>trans</i> fats,<br>weight gain, anorexia<br>nervosa | Weight gain, very-low-fat<br>diets, high intake<br>of refined carbohydrates,<br>excessive alcohol intake |
| Drugs | Diuretics, cyclosporine,<br>glucocorticoids,<br>amiodarone | Oral estrogens, glucocorticoids, bile acid sequestrants, protease inhibitors, retinoic acid, anabolic steroids, sirolimus, raloxifene, tamoxifen, beta blockers (not carvedilol), thiazides |
| Diseases | Biliary obstruction,<br>nephrotic syndrome | Nephrotic syndrome,<br>chronic renal failure,<br>lipodystrophies |
| Disorders and altered states of metabolism | Hypothyroidism,<br>obesity, pregnancy* | Diabetes (poorly controlled),<br>hypothyroidism, obesity;<br>pregnancy* |

Adapted with permission from Stone et al (80).

<sup>\*</sup>Fasting lipid panel preferred. In a nonfasting individual, a non-HDL-C level  $\geq$ 220 mg/dL could indicate genetic hypercholesterolemia that requires further evaluation or a secondary etiology. If nonfasting triglycerides are  $\geq$ 500 mg/dL, a fasting lipid panel is required.

<sup>†</sup>It is reasonable to evaluate the potential for ASCVD benefits and for adverse effects, and to consider patient preferences, in initiating or continuing a moderate- or high-intensity statin in individuals with ASCVD who are >75 years of age.

<sup>\*</sup>Cholesterol and triglycerides rise progressively throughout pregnancy (80); treatment with statins, niacin, and ezetimibe are contraindicated during pregnancy and lactation. LDL-C indicates low-density lipoprotein cholesterol.



Figure 4. Initiating Statin Therapy in Individuals Without Clinical ASCVD

Colors correspond to the Classes of Recommendation in Table 1.

\*Fasting lipid panel preferred. In a nonfasting individual, a non-HDL-C level ≥220 mg/dL could indicate genetic hypercholesterolemia that requires further evaluation or a secondary etiology. If nonfasting triglycerides are ≥500 mg/dL, a fasting lipid panel is required.

†The Pooled Cohort Equations can be used to estimate 10-year ASCVD risk in individuals with and without diabetes.

A downloadable spreadsheet enabling estimation of 10-year and lifetime risk for ASCVD and a Web-based calculator are available at http://my.americanheart.org/cvriskcalculator and http://www.cardiosource.org/en/Science-And-Quality/Practice-Guidelines-and-Quality-Standards/2013-Prevention-Guideline-Tools.aspx.

 $\ddagger$ For those in whom a risk assessment is uncertain, consider factors such as primary LDL-C  $\ge$ 160 mg/dL or other evidence of genetic hyperlipidemias; family history of premature ASCVD with onset <55 years of age in a first-degree male relative or <65 years of age in a first-degree female relative, high-sensitivity C-reactive protein  $\ge$ 2 mg/L; CAC  $\ge$ 300 Agaston units or  $\ge$ 75th percentile for age, sex, and ethnicity (for additional information, see http://www.mesa-nhlbi.org/CACReference.aspx); ABI <0.9; or lifetime risk of ASCVD. Additional factors that may aid in individual risk assessment could be identified in the future.

§1) Potential ASCVD risk-reduction benefits. The absolute reduction in ASCVD events from moderate- or high-intensity statin therapy can be approximated by multiplying the estimated 10-year ASCVD risk by the anticipated relative-risk reduction from the intensity of statin initiated (~30% for moderate-intensity statin or ~45% for high-intensity statin therapy). The net ASCVD risk-reduction benefit is estimated from the number of potential ASCVD events prevented with a statin, compared to the number of potential excess adverse effects. 2) Potential adverse effects. The excess risk of diabetes is the main consideration in ~0.1 excess cases per 100 individuals treated with a moderate-intensity statin for 1 year and ~0.3 excess cases per 100 individuals treated with a high-intensity statin for 1 year. In RCTs, both statin-treated and placebo-treated participants experienced the same rate of muscle symptoms. The actual rate of statin-related muscle symptoms in the clinical population is unclear. Muscle symptoms attributed to statin therapy should be evaluated (see Table 8, Safety Recommendation 8).

ABI indicates ankle-brachial index; ALT, alanine transaminase; ASCVD, atherosclerotic cardiovascular disease; CAC, coronary artery calcium; CK, creatine kinase; FH, familial hypercholesterolemia; LDL-C, low-density lipoprotein cholesterol; MI, myocardial infarction; RCT, randomized controlled trial; and ULN, upper limit of normal.

of other risk factors to reduce their ASCVD event rates. Therefore, it is reasonable to use high-intensity statin therapy to achieve at least a 50% reduction. It is recognized that maximal statin therapy might not be adequate to lower LDL-C sufficiently to reduce ASCVD event risk in individuals with primary severe elevations of LDL-C. In addition to a maximally tolerated dose of statin, nonstatin cholesterol-lowering medications are often needed to lower LDL-C to acceptable levels in these individuals. Because the hypercholesterolemia in these high-risk individuals is often genetically determined, family screening is especially important in this group to identify additional family members who would benefit from assessment and early treatment.

Secondary causes of severe elevations of LDL-C ≥190 mg/dL and triglycerides ≥500 mg/dL often contribute to the magnitude of the hyperlipidemia and should be evaluated and treated appropriately. For guidance, we note that in a lipid specialty clinic, the most frequently encountered secondary conditions were excessive alcohol intake, uncontrolled diabetes, and overt albuminuria (79). Table 6 focuses on secondary causes of hyperlipidemia most likely encountered in clinical practice (80). Management of individuals with fasting triglycerides ≥500 mg/dL has been addressed in an AHA statement (45).

The flow diagram for the initiation and management of statin therapy in individuals with LDL-C  $\geq$ 190 mg/dL is provided in Figure 4.

### 4.5. Primary Prevention in Individuals With Diabetes

A high level of evidence supports the use of moderateintensity statin therapy in persons with diabetes who are 40 to 75 years of age. The only trial of high-intensity statin therapy in primary prevention was performed in a population without diabetes. However, a high level of evidence existed for event reduction with statin therapy in individuals with a  $\geq$ 7.5% estimated 10-year ASCVD risk (Section 4.6) who did not have diabetes to recommend high-intensity statin therapy preferentially for individuals with diabetes and a  $\geq$ 7.5% estimated 10-year ASCVD risk (Section 4.7). This consideration for those with diabetes who are 40 to 75 years of age recognizes that these individuals are at substantially increased lifetime risk for ASCVD events and death. Moreover, individuals with diabetes experience greater morbidity and worse survival after the onset of clinical ASCVD. In persons with diabetes who are <40 years of age or >75 years of age, or whose LDL-C is <70 mg/dL, statin therapy should be individualized on the basis of considerations of ASCVD risk-reduction benefits, the potential for adverse effects and drug-drug interactions, and patient preferences (Figure 4).

### 4.6. Primary Prevention in Individuals Without Diabetes and With LDL-C 70 to 189 mg/dL

In individuals 40 to 75 years of age with LDL-C 70 to 189 mg/dL who do not have clinical ASCVD or diabetes,

### Table 7. Rationale for the Expert Panel Approach to Primary-Prevention Guidelines

- Cholesterol-lowering medications, particularly statins, are efficacious and effective for reducing risk of initial cardiovascular events.
- Statins are associated with similar relative risk reductions for cardiovascular events across the majority of primary-prevention patient groups studied.\*
- The extent of relative risk reduction for ASCVD is proportional to the degree of LDL-C lowering observed on statin therapy. Therefore, more intensive statin therapy could reduce risk more than moderate- or lower-intensity statin therapy.
- According to consistent findings, the absolute benefit in ASCVD risk reduction is proportional to the baseline risk of the patient group or individual and to the intensity of statin therapy.
- Patients or groups at higher baseline absolute risk, therefore, will derive greater absolute benefit from initiation of statin therapy over a period of 5 to 10 years.
- 6. The absolute risk for adverse outcomes, including a small excess in cases of newly diagnosed diabetes, also appears to be proportional to the intensity of statin therapy. However, the adverse outcome of incident (or earlier diagnosis of) diabetes must be weighed in the context of the potentially fatal or debilitating occurrence of MI or stroke that could be prevented by statin therapy.
- 7. The Expert Panel emphasizes that the occurrence of a major ASCVD event (MI or stroke) represents a much greater harm to health status than does an increase in blood glucose leading to a diagnosis of diabetes. The net absolute benefit of statin therapy can be considered as a comparison of the absolute risk reduction for ASCVD with the absolute excess risks, including that for diabetes. Benefit also could be understood as a comparison of the number of statin-treated patients that would result in the prevention of 1 case of major ASCVD (NNT) with the number of statin-treated patients that would result in 1 excess case of diabetes (NNH).
- 8. Because the absolute benefit in terms of ASCVD risk reduction depends on the baseline absolute risk for ASCVD, the absolute benefit from initiation of statin therapy is lower and would approach the risk for adverse effects in patients with lower baseline levels of predicted ASCVD risk.
- Available RCT evidence indicates a clear net absolute benefit of initiation of moderate-to-intensive statin therapy at a baseline estimated 10-year ASCVD risk of ≥7.5%.
- 10. Available RCT evidence indicates that when baseline ASCVD risk is 5.0% to <7.5%, there is still net absolute benefit with moderate-intensity statin therapy. However, the tradeoffs between the ASCVD risk-reduction benefit and adverse effects are less clear. Thus, a clinician-patient discussion is even more important for individuals with this range of ASCVD risk. The net benefit of high-intensity statin therapy may be marginal in such individuals.</p>

#### Conclusion

On the basis of the above tenets and its review of the evidence, this guideline recommends initiation of moderate or intensive statin therapy for patients who are eligible for primary ASCVD prevention and have a predicted 10-year "hard" ASCVD risk of  $\geq\!7.5\%$ . This guideline recommends that initiation of moderate-intensity statin therapy be considered for patients with predicted 10-year "hard" ASCVD risk of 5.0% to  $<\!7.5\%$ .

ASCVD indicates atherosclerotic cardiovascular disease; CVD, cardiovascular disease; LDL-C, low-density lipoprotein cholesterol; MI, myocardial infarction; NNH, number needed to harm; NNT, number needed to treat; NYHA, New York Heart Association; and RCT, randomized controlled trial.

<sup>\*</sup>Available evidence suggests that initiation of statin therapy might not achieve a significant reduction of CVD risk in patients with higher classes of NYHA heart failure or who are receiving maintenance hemodialysis.

initiation of statin therapy based on estimated 10-year ASCVD risk is recommended, regardless of sex, race, or ethnicity (Section 4.7). Point estimates of statin-associated reductions in the relative risk of ASCVD in primary prevention are similar for both women and men. There also is no evidence that the ASCVD risk-reduction benefit or adverse-effect profiles differ by race.

To better identify those individuals without ASCVD who would most benefit from statin therapy to reduce ASCVD risk, data were used from the 3 exclusively primary-prevention RCTs that included individuals with LDL-C levels <190 mg/dL, almost all of whom had LDL-C levels  $\geq 70 \text{ mg/dL } (17,18,49)$ . From these trials, an estimate of the expected 10-year ASCVD event rates was derived from the placebo groups. The rates of excess adverse events in the statin treatment groups were obtained from meta-analyses of statin RCTs. A high level of evidence for an ASCVD risk-reduction benefit from initiation of moderate- or high-intensity statin therapy in individuals 40 to 75 years of age with  $\geq$ 7.5% estimated 10year ASCVD risk was found (Section 4.7). The reduction in ASCVD risk clearly outweighs the potential for adverse effects (Table 7). Thus, it is recommended that individuals 40 to 75 years of age, who are not already candidates for statin therapy on the basis of the presence of clinical ASCVD, diabetes, or LDL-C  $\geq$ 190 mg/dL, receive statin therapy if they have a  $\geq 7.5\%$  estimated 10-year risk for ASCVD and LDL-C 70 to 189 mg/dL. Although only 1 exclusively primary-prevention RCT included individuals with LDL-C 70 to <100 mg/dL, the Cholesterol Treatment Trialists 2010 meta-analysis found a relative reduction in ASCVD events of similar magnitude across the spectrum of LDL-C levels  $\geq$ 70 mg/dL (20). Given that the relative risk reduction is similar across the range of LDL-C 70 to 189 mg/dL, the absolute benefit of statin therapy in primary prevention is determined by the global risk estimate using all the risk factor information and is reflected in the estimated 10-year ASCVD risk.

A conservative estimate of adverse events includes excess cases of new-onset diabetes and rare cases of myopathy and hemorrhagic stroke. The rate of excess diabetes varies by statin intensity. For moderate-intensity statins, approximately 0.1 excess case of diabetes per 100 statin-treated individuals per year has been observed, and for high-intensity statins, approximately 0.3 excess case of diabetes per 100 statin-treated individuals per year has been observed (52,81). The long-term adverse effects of statin-associated cases of diabetes over a 10-year period are unclear and are unlikely to be equivalent to an MI, stroke, or ASCVD death. Myopathy (~0.01 excess case per 100) and hemorrhagic stroke (~0.01 excess case per 100) make minimal contributions to excess risk from statin therapy (13).

Although a similar level of evidence of a reduction in ASCVD events from moderate- and high-intensity statin therapy is present for those with a 5% to <7.5% estimated 10-year ASCVD risk, the potential for adverse effects may

outweigh the potential for ASCVD risk-reduction benefit when high-intensity statin therapy is used in this risk group. However, for moderate-intensity statin therapy, the ASCVD risk reduction clearly exceeds the potential for adverse effects.

Before initiating statin therapy for the primary prevention of ASCVD in adults with  $\geq$ 7.5% or 5% to <7.5% estimated 10-year ASCVD risk, it is reasonable for clinicians and patients to engage in a discussion of the proposed therapy. This discussion should include the potential for ASCVD benefit, the potential for adverse effects and drug-drug interactions, and consideration of patient preferences for treatment.

No primary-prevention RCT data were available for individuals 21 to 39 years of age, and few data were available for individuals >75 years of age. Additionally, in individuals 40 to 75 years of age with <5% estimated 10year ASCVD risk, the net benefit from statin therapy over a 10-year period may be small. Therefore, in adults with LDL-C <190 mg/dL who are not otherwise identified in a statin benefit group or for whom a risk-based treatment decision is uncertain after quantitative risk assessment, clinician knowledge, experience, and skill ("the art of medicine") and patient preferences all contribute to the decision to initiate statin therapy (82). Before initiation of statin therapy, the clinician-patient discussion should include consideration of the potential for ASCVD riskreduction benefits, adverse effects, and drug-drug interactions. Additional factors may also be considered to inform treatment decision making in selected individuals. Factors that can contribute to assessment of ASCVD risk include primary LDL-C ≥160 mg/dL or other evidence of genetic hyperlipidemias; family history of premature ASCVD with onset <55 years of age in a first-degree male relative or <65 years of age in a first-degree female relative; high-sensitivity C-reactive protein >2 mg/L, coronary artery calcium score ≥300 Agatston units or ≥75th percentile for age, sex, and ethnicity (for additional information, see http://www.mesa-nhlbi.org/CACReference.aspx); ankle-brachial index <0.9; or elevated lifetime risk of ASCVD. Additional factors that might aid in individual risk assessment could be identified in the future.

For an individual <40 years of age, the 10-year horizon might not be optimal for predicting lifetime risk of ASCVD (see 2013 ACC/AHA Guideline on the Assessment of Cardiovascular Risk) (11). Future RCTs will be needed to determine the optimal age at which to initiate statin therapy to reduce ASCVD risk, as well as to determine the optimum duration of statin therapy.

#### 4.7. Risk Assessment in Primary Prevention

To estimate more closely the total burden of ASCVD, this guideline recommends a comprehensive assessment of the estimated 10-year risk for an ASCVD event that includes both CHD and stroke. This is in contrast to the use of an estimated 10-year risk for hard CHD (defined as nonfatal MI and CHD death) (83).

This guideline recommends using the new Pooled Cohort Risk Assessment Equations developed by the Risk Assessment Work Group to estimate the 10-year ASCVD risk (defined as first-occurrence nonfatal and fatal MI and nonfatal and fatal stroke) for the identification of candidates for statin therapy (see http://my.americanheart.org/ cvriskcalculator and http://www.cardiosource.org/en/ Science-And-Quality/Practice-Guidelines-and-Quality-Standards/2013-Prevention-Guideline-Tools.aspx for risk calculator). These equations should be used to predict stroke as well as CHD events in non-Hispanic, Caucasian, and African-American women and men 40 to 79 years of age with or without diabetes who have LDL-C levels 70 to 189 mg/dL and are not receiving statin therapy. A more complete discussion of risk assessment is provided in the Full Panel Report Supplement.

This guideline does not require specific risk factor counting for risk assessment or the use of RCT risk factor inclusion criteria to determine statin eligibility. Rather, a global ASCVD risk assessment to guide initiation of statin therapy was chosen for several important reasons (see rationale in Table 7 and further discussion in Section 7.3 of the Full Panel Report Supplement): 1) The Cholesterol Treatment Trialists individual-level meta-analyses were used to evaluate the effect of statins in various important patient subgroups, including risk factor cutpoints used for RCT eligibility. The Expert Panel found that statin therapy reduces ASCVD events regardless of risk factor characteristics in both primary and secondary prevention. Therefore, the rationale for using fixed cutpoints to determine whether statin therapy should be used is refuted by a consideration of the total body of evidence. 2) Use of absolute ASCVD risk facilitates a quantitative assessment of the potential for an ASCVD risk-reduction benefit as compared with the potential for adverse effects. 3) Use of an RCT eligibility criteria-based approach results in failure to identify a substantial proportion of higher-risk individuals who could benefit from statin therapy and overidentification of very-low-risk individuals who might not experience a net benefit from statin therapy over a 10-year period.

#### 4.8. Heart Failure and Hemodialysis

No recommendation was made with regard to the initiation or continuation of statin therapy in 2 specific groups: 1) individuals with New York Heart Association class II—IV heart failure, and 2) individuals undergoing maintenance hemodialysis. In the 4 RCTs reviewed that specifically addressed statin treatment in these groups, there were individuals with and without heart disease (84–87). Although statin therapy did not reduce ASCVD events in 2 RCTs for each condition (84–87), there was insufficient information on which to base recommendations for or against statin treatment. Future research may identify subgroups of patients with these conditions that may benefit from statin therapy. In individuals with these

conditions, the potential for ASCVD risk-reduction benefits, adverse effects, and drug-drug interactions, along with other cautions and contraindications to statin therapy and choice of statin dose, must also be considered by the treating clinician.

#### 5. Safety: Recommendations

See safety recommendations for statins (Table 8) and nonstatin drugs (Table 9).

RCT data were also used to examine the safety of lipid medications. From the statin RCTs and meta-analyses, patient characteristics and monitoring strategies were identified that should enhance the safe use of high- and moderate-intensity statin therapy. Patient characteristics that may influence statin safety include but are not limited to: multiple or serious comorbidities, including impaired renal or hepatic function; a history of previous statin intolerance or muscle disorders; concomitant use of drugs affecting statin metabolism; a history of hemorrhagic stroke; and age >75 years. Asian ancestry may also influence the initial choice of statin intensity.

This guideline recommends against routine measurement of creatine kinase in individuals receiving statin therapy. This measurement should be reserved for those with muscle symptoms. However, measurement of a baseline creatine kinase may be useful in those at increased risk of adverse muscle events. Such individuals include those with a personal or family history of statin intolerance or muscle disease, clinical presentation, or concomitant drug therapy that might increase the likelihood of myopathy.

Expert recommendations are also provided for managing muscle symptoms while a patient is on statin therapy. These useful management suggestions were derived from other clinical trial data and clinical experience to enhance the safety and tolerability of statin therapy. Consistent with the protocols of the RCTs, patients should be asked at each visit, both before and after initiation of statin therapy, about muscle symptoms such as muscle weakness or fatigue, aching, pain, tenderness, cramps, or stiffness. The recommended approach for management of muscle symptoms is described in Table 8, Recommendation 8.

This guideline recommends that baseline measurement of transaminase (alanine transaminase; ALT) levels should be performed before initiation of statin therapy. This approach was taken in the RCTs reviewed for this report. There is no recommendation to monitor transaminase (ALT) levels because ALT monitoring was performed in the RCTs, and there was no significant difference between placebo groups and statin treatment groups in the rates of ALT elevations. In addition, the U.S. Food and Drug Administration has indicated that if the baseline hepatic transaminases are normal, further hepatic monitoring is not needed. During statin therapy, it is reasonable to measure hepatic function if symptoms suggesting

**Table 8. Statin Safety Recommendations** 

| Recommendations | NHLBI Grade | NHLBI Evidence<br>Statements | ACC/AHA COR | ACC/AHA LOE |
|---|---|---|---|---|
| Safety | | | | |
| To maximize the safety of statins, selection of the appropriate statin and dose in men and nonpregnant/nonnursing women should be based on patient characteristics, level of ASCVD* risk, and potential for adverse effects. Moderate-intensity statin therapy should be used in individuals in whom high-intensity statin therapy would otherwise be recommended when characteristics predisposing them to statin-associated adverse effects are | A (Strong) | 46-55 | ' | В |
| present. Characteristics predisposing individuals to statin adverse effects include but are not limited to: | | | | |
| Multiple or serious comorbidities, including impaired renal or hepatic function. | | | | |
| <ul> <li>History of previous statin intolerance or muscle disorders.</li> </ul> | | | | |
| <ul> <li>Unexplained ALT elevations ≥3 times ULN.</li> </ul> | | | | |
| <ul> <li>Patient characteristics or concomitant use of drugs affecting statin<br/>metabolism.</li> <li>Age &gt;75 years.</li> </ul> | | | | |
| Additional characteristics that could modify the decision to use higher statin intensities might include but are not limited to: | | | | |
| History of hemorrhagic stroke. | | | | |
| Asian ancestry. | | | | |
| 2a. CK should not be routinely measured in individuals receiving statin therapy. | A (Strong) | 45,49-51,54,55 | III: No Benefit | A |
| 2b. Baseline measurement of CK is reasonable for individuals believed to be at increased risk for adverse muscle events because of a personal or family history of statin intolerance or muscle disease, clinical presentation, or concomitant drug therapy that might increase the risk of myopathy. | E (Expert Opinion) | _ | lla | <b>C</b> (88) |
| During statin therapy, it is reasonable to measure CK in individuals with muscle symptoms, including pain, tenderness, stiffness, cramping, weakness, or generalized fatigue. | E (Expert Opinion) | _ | lla | <b>C</b> (88) |
| 3a. Baseline measurement of hepatic transaminase levels (ALT) should be performed before initiation of statin therapy. | B (Moderate) | 46,52,53 | I† | В |
| 3b. During statin therapy, it is reasonable to measure hepatic function if<br>symptoms suggesting hepatotoxicity arise (e.g., unusual fatigue or weakness,<br>loss of appetite, abdominal pain, dark-colored urine, or yellowing of the skin<br>or sclera). | E (Expert Opinion) | _ | lla | <b>C</b> (89) |
| <ol> <li>Decreasing the statin dose may be considered when 2 consecutive values<br/>of LDL-C levels are &lt; 40 mg/dL.</li> </ol> | C (Weak) | 45 | llb | С |
| 5. It may be harmful to initiate simvastatin at 80 mg daily or increase the dose of simvastatin to 80 mg daily. | B (Moderate) | 6,54 | III: Harm | <b>A</b><br>(67,90) |
| 6. Individuals receiving statin therapy should be evaluated for new-onset diabetes according to the current diabetes screening guidelines (91). Those who develop diabetes during statin therapy should be encouraged to adhere to a heart-healthy dietary pattern, engage in physical activity, achieve and maintain a healthy body weight, cease tobacco use, and continue statin therapy to reduce their risk of ASCVD events. | B (Moderate) | 44 | I‡ | В |
| 7. For individuals taking any dose of statins, it is reasonable to use caution in individuals >75 years of age, as well as in individuals who are taking concomitant medications that alter drug metabolism, taking multiple drugs, or taking drugs for conditions that require complex medication regimens (e.g., those who have undergone solid organ transplantation or are receiving treatment for HIV). A review of the manufacturer's prescribing information may be useful before initiation of any cholesterol-lowering drug. | E (Expert Opinion) | _ | lla | <b>C</b><br>(16,64-70,<br>89,92-94) |

Continued on the next page

hepatotoxicity arise (e.g., unusual fatigue or weakness, loss of appetite, abdominal pain, dark-colored urine, or yellowing of the skin or sclera).

Decreasing the statin dose may be considered when 2 consecutive values of LDL-C are <40 mg/dL. This recommendation was based on the approach taken in 2 RCTs. However, no data were identified that suggest an excess of adverse events occurred when LDL-C levels were below this level.

Statins modestly increase the excess risk of type 2 diabetes in individuals with risk factors for diabetes. The potential for an ASCVD risk-reduction benefit outweighs the excess risk of diabetes in all but the lowest-risk individuals (Section 4.5). All individuals receiving statins should be counseled on healthy-lifestyle habits. Individuals receiving statin therapy should be evaluated for new-onset diabetes according to the current diabetes screening guidelines (91). Those who develop diabetes

**Table 8. Continued** 

9.

| ecommendations | NHLBI Grade | NHLBI Evidence<br>Statements | ACC/AHA COR | ACC/AHA LOE |
|---|---|---|---|---|
| <ul> <li>It is reasonable to evaluate and treat muscle symptoms, including pain, tenderness, stiffness, cramping, weakness, or fatigue, in statin-treated patients according to the following management algorithm:</li> <li>To avoid unnecessary discontinuation of statins, obtain a history of prior or current muscle symptoms to establish a baseline before initiation of statin therapy.</li> <li>If unexplained severe muscle symptoms or fatigue develop during statin therapy, promptly discontinue the statin and address the possibility of rhabdomyolysis by evaluating CK and creatinine and performing urinalysis for myoglobinuria.</li> <li>If mild to moderate muscle symptoms develop during statin therapy: <ul> <li>Discontinue the statin until the symptoms can be evaluated.</li> <li>Evaluate the patient for other conditions that might increase the risk for muscle symptoms (e.g., hypothyroidism, reduced renal or hepatic function, rheumatologic disorders such as polymyalgia rheumatica, steroid myopathy, vitamin D deficiency, or primary muscle diseases).</li> <li>If muscle symptoms resolve, and if no contraindication exists, give the patient the original or a lower dose of the same statin to establish a causal relationship between the muscle symptoms and statin therapy.</li> <li>If a causal relationship exists, discontinue the original statin. Once muscle symptoms resolve, use a low dose of a different statin.</li> <li>Once a low dose of a statin is tolerated, gradually increase the dose as tolerated.</li> <li>If, after 2 months without statin treatment, muscle symptoms or elevated CK levels do not resolve completely, consider other causes of muscle symptoms listed above.</li> <li>If persistent muscle symptoms are determined to arise from a condition unrelated to statin therapy, or if the predisposing condition has been treated, resume statin therapy at the original dose.</li> </ul> </li> </ul> | E (Expert Opinion) | | lla | B<br>(15,88,96-98) |
| For individuals presenting with a confusional state or memory impairment<br>while on statin therapy, it may be reasonable to evaluate the patient for<br>nonstatin causes, such as exposure to other drugs, as well as for systemic and<br>neuropsychiatric causes, in addition to the possibility of adverse effects<br>associated with statin drug therapy. | E (Expert Opinion) | _ | IIb | <b>C</b> (38,89,99,100) |

<sup>\*</sup>Based on the presence of clinical ASCVD, diabetes, LDL-C >190 mg/dL, or level of estimated 10-year ASCVD risk.

 $\dagger$ Individuals with elevated ALT levels (usually >1.5 or 2 times ULN) were excluded from RCT participation. Unexplained ALT  $\geq$ 3 times ULN is a contraindication to statin therapy as listed in manufacturer's prescribing information.

Statin use is associated with a very modest excess risk of new-onset diabetes in RCTs and meta-analyses of RCTs (i.e., ~0.1 excess cases per 100 individuals treated for 1 year with moderate-intensity statin therapy and ~0.3 excess cases per 100 individuals treated for 1 year with high-intensity statin therapy. The increased risk of new-onset diabetes appears to be confined to those with risk factors for diabetes. These individuals are also at higher risk of ASCVD because of these risk factors. Therefore, if a statin-treated individual develops diabetes as detected by current diabetes screening guidelines, he or she should be counseled to adhere to a heart-healthy dietary pattern, engage in physical activity, achieve and maintain a healthy body weight, cease tobacco use, and continue statin therapy to reduce the risk of ASCVD events.

ACC indicates American College of Cardiology; AHA, American Heart Association; ALT, alanine transaminase; ASCVD, atherosclerotic cardiovascular disease; CK, creatine kinase; COR, Class of Recommendation; NHLBI, National Heart, Lung, and Blood Institute; LDL-C, low-density lipoprotein cholesterol; LOE, Level of Evidence; RCTs, randomized controlled trials; ULN, upper limit of normal; and —, not applicable.

during statin therapy should be encouraged to adhere to a heart-healthy dietary pattern, engage in physical activity, achieve and maintain a healthy body weight, cease tobacco use, and continue statin therapy to reduce their risk of ASCVD events.

Statins are listed as pregnancy category X and should not be used in women of childbearing potential unless these women are using effective contraception and are not nursing.

For individuals taking any dose of statins, it is reasonable to use caution in individuals >75 years of age, as well as in individuals who are taking concomitant medications that alter drug metabolism, taking multiple drugs, or taking drugs for conditions that require complex medication regimens (e.g., those who have undergone solid

organ transplantation or are receiving treatment for HIV). A review of the manufacturer's prescribing information might be useful before initiation of any cholesterol-lowering drug, because RCTs considered defined populations and many patients in everyday practice would not qualify for clinical trials. Thus, clinicians should also consult other sources of safety data, such as pharmacists, drug information centers, and manufacturers' prescribing information on a regular basis for up-to-date guidance about lipid medications and medication interactions.

Statins used in combination with other cholesterollowering drug therapies might require more intensive monitoring. The safety of nonstatin agents was reviewed, and that information is included in Table 9 and the Full Panel Report Supplement. Warnings about the use of

**Table 9. Nonstatin Safety Recommendations** 

| Recommendations | NHLBI Grade | NHLBI Evidence<br>Statements | ACC/AHA COR | ACC/AHA LOE |
|---|---|---|---|---|
| Safety of Niacin 1. Baseline hepatic transaminases, fasting blood glucose or hemoglobin A1c, and uric acid should be obtained before initiation of niacin, and again during up-titration to a maintenance dose and every 6 months thereafter. | B (Moderate) | 77 | 1 | В |
| 2. Niacin should not be used if: | | | | |
| Hepatic transaminase elevations are higher than 2 to 3 times ULN. | A (Strong) | 79 | III: Harm | В - |
| <ul> <li>Persistent severe cutaneous symptoms, persistent hyperglycemia, acute<br/>gout, or unexplained abdominal pain or gastrointestinal symptoms occur.</li> </ul> | B (Moderate) | 78,79 | III: Harm | В |
| New-onset atrial fibrillation or weight loss occurs. | C (Weak) | 80 | III: Harm | B<br>B |
| <ol><li>In individuals with adverse effects from niacin, the potential for ASCVD<br/>benefits and the potential for adverse effects should be reconsidered before<br/>reinitiation of niacin therapy.</li></ol> | E (Expert) | _ | · | (9,101-104) |
| 4. To reduce the frequency and severity of adverse cutaneous symptoms, it is<br>reasonable to: | E (Expert) | _ | lla | <b>C</b><br>(9,101-104) |
| <ul> <li>Start niacin at a low dose and titrate to a higher dose over a period of weeks as tolerated.</li> <li>Take niacin with food or premedicate with aspirin 325 mg 30 minutes before niacin dosing to alleviate flushing symptoms.</li> </ul> | | | | |
| <ul> <li>If an extended-release preparation is used, increase the dose of extended-release niacin from 500 mg to a maximum of 2,000 mg/day over 4 to 8 weeks, with the dose of extended-release niacin increasing not more than weekly.</li> </ul> | | | | |
| <ul> <li>If immediate-release niacin is chosen, start at a dose of 100 mg 3 times<br/>daily and up-titrate to 3 g/day, divided into 2 or 3 doses.</li> </ul> | | | | |
| Safety of BAS | | | | |
| <ol> <li>BAS should not be used in individuals with baseline fasting triglyceride<br/>levels ≥300 mg/dL or type III hyperlipoproteinemia, because severe<br/>triglyceride elevations might occur. (A fasting lipid panel should be obtained<br/>before BAS is initiated, 3 months after initiation, and every 6 to 12 months<br/>thereafter.)</li> </ol> | C (Weak) | 60 | III: Harm | В |
| <ol> <li>It is reasonable to use BAS with caution if baseline triglyceride levels are<br/>250 to 299 mg/dL, and evaluate a fasting lipid panel in 4 to 6 weeks after<br/>initiation. Discontinue the BAS if triglycerides exceed 400 mg/dL.</li> </ol> | E (Expert) | _ | lla | <b>C</b> (105) |
| Safety of Cholesterol-Absorption Inhibitors | | | | |
| <ol> <li>It is reasonable to obtain baseline hepatic transaminases before initiation of<br/>ezetimibe. When ezetimibe is coadministered with a statin, monitor trans-<br/>aminase levels as clinically indicated, and discontinue ezetimibe if persistent<br/>ALT elevations ≥3 times ULN occur.</li> </ol> | C (Weak) | 61-64 | lla | В |
| Safety of Fibrates | | | | _ |
| <ol> <li>Gemfibrozil should not be initiated in patients on statin therapy because of an<br/>increased risk for muscle symptoms and rhabdomyolysis.</li> </ol> | B (Moderate) | 46 | III: Harm | В |
| <ol><li>Fenofibrate may be considered concomitantly with a low- or moderate-<br/>intensity statin only if the benefits from ASCVD risk reduction or triglyceride<br/>lowering when triglycerides are ≥500 mg/dL are judged to outweigh the<br/>potential risk for adverse effects.</li></ol> | E (Expert) | _ | IIb | <b>C</b><br>(14) |
| 3. Renal status should be evaluated before fenofibrate initiation, within 3 months after initiation, and every 6 months thereafter. Assess renal safety with both a serum creatinine level and an eGFR based on creatinine. | B (Moderate) | 66,67 | - 1 | В |
| <ul> <li>Fenofibrate should not be used if moderate or severe renal impairment, defined as eGFR &lt;30 mL/min per 1.73 m², is present.</li> <li>If eGFR is between 30 and 59 mL/min per 1.73 m², the dose of fenofibrate should not exceed 54 mg/day.*</li> <li>If, during follow-up, the eGFR decreases persistently to ≤30 mL/min per 1.73 m², fenofibrate should be discontinued.</li> </ul> | | | III: Harm | В |
| Safety of Omega-3 Fatty Acids 1. If EPA and/or DHA are used for the management of severe hypertriglyceridemia, defined as triglycerides ≥500 mg/dL, it is reasonable to evaluate the patient for gastrointestinal disturbances, skin changes, and bleeding. | C (Weak) | 70 | lla | В |

<sup>\*</sup>Consult the manufacturer's prescribing information as there are several forms of fenofibrate available.

ACC indicates American College of Cardiology; AHA, American Heart Association; ALT, alanine transaminase; ASCVD, atherosclerotic cardiovascular disease; BAS, bile acid sequestrants; COR, Class of Recommendation; DHA, docosahexanoic acid; EPA, eicosapentaenoic acid; eGFR, estimated glomerular filtration rate; LOE, Level of Evidence; NHLBI, National Heart, Lung, and Blood Institute; ULN, upper limit of normal; and —, not applicable.

Table 10. Recommendations for Monitoring, Optimizing, and Addressing Insufficient Response to Statin Therapy

| Recommendations | NHLBI Grade | NHLBI Evidence<br>Statements | ACC/AHA COR | ACC/AHA LOE |
|---|---|---|---|---|
| Monitoring Statin Therapy 1. Adherence to medication and lifestyle, therapeutic response to statin therapy, and safety should be regularly assessed. This should also include a fasting lipid panel performed within 4-12 weeks after initiation or dose adjustment, and every 3-12 months thereafter. Other safety measurements should be measured as clinically indicated. | A (Strong) | 45 | 1 | A |
| Optimizing Statin Therapy | | | | |
| <ol> <li>The maximum tolerated intensity of statin should be used in individuals for<br/>whom a high- or moderate-intensity statin is recommended but not tolerated.</li> </ol> | B (Moderate) | 25,26,27,45 | <b>[</b> * | В |
| Insufficient Response to Statin Therapy | | | | |
| <ol> <li>In individuals who have a less-than-anticipated therapeutic response or are intolerant of the recommended intensity of statin therapy, the following should be performed: <ul> <li>Reinforce medication adherence.</li> <li>Reinforce adherence to intensive lifestyle changes.</li> <li>Exclude secondary causes of hyperlipidemia.</li> </ul> </li> </ol> | A (Strong) | 45 | 1 | A |
| <ul> <li>2. It is reasonable to use the following as indicators of anticipated therapeutic response to the recommended intensity of statin therapy. Focus is on the intensity of the statin therapy. As an aid to monitoring: <ul> <li>High-intensity statin therapy† generally results in an average LDL-C reduction of ≥50% from the untreated baseline.</li> <li>Moderate-intensity statin therapy generally results in an average LDL-C reduction of 30% to &lt;50% from the untreated baseline.</li> <li>LDL-C levels and percents reduction are to be used only to assess response to therapy and adherence. They are not to be used as performance standards.</li> </ul> </li> </ul> | E (Expert Opinion) | _ | lla | B<br>(46-48,78,<br>106,107) |
| 3. In individuals at higher ASCVD risk receiving the maximum tolerated intensity of statin therapy who continue to have a less-than-anticipated therapeutic response, addition of nonstatin cholesterol-lowering drug(s) may be considered if the ASCVD risk-reduction benefits outweigh the potential for adverse effects. Higher-risk individuals include: Individuals with clinical ASCVD‡ <75 years of age. Individuals with baseline LDL-C ≥190 mg/dL. Individuals 40-75 years of age with diabetes. Preference should be given to nonstatin cholesterol-lowering drugs shown to reduce ASCVD events in RCTs. | E (Expert Opinion) | _ | lib | C<br>(9,14,108-110) |
| 4. In individuals who are candidates for statin treatment but are completely<br>statin intolerant, it is reasonable to use nonstatin cholesterol-lowering drugs<br>that have been shown to reduce ASCVD events in RCTs if the ASCVD risk-<br>reduction benefits outweigh the potential for adverse effects. | E (Expert Opinion) | _ | lla | <b>B</b> (88,101,111-116) |

<sup>\*</sup>Several RCTs found that low-intensity and low-moderate-intensity statin therapy reduced ASCVD events. In addition, the Cholesterol Treatment Trialists meta-analyses found that each 39-mg/dL reduction in LDL-C reduces ASCVD risk by 22%. Therefore, the Panel considered that submaximal statin therapy should be used to reduce ASCVD risk in those unable to tolerate moderate- or high-intensity statin therapy.

cholesterol-lowering agents in pregnancy and lactation also apply to nonstatins, and the manufacturer's prescribing information should be consulted.

### 6. Managing Statin Therapy: Recommendations

See Table 10 for a summary of recommendations for monitoring, optimizing, and addressing insufficient response to statin therapy.

#### **6.1.** Monitoring Statin Therapy

A high level of RCT evidence supports the use of an initial fasting lipid panel (total cholesterol, triglycerides, HDL-C, and calculated LDL-C), followed by a second lipid panel 4 to 12 weeks after initiation of statin therapy, to determine a patient's adherence. Thereafter, assessments should be performed every 3 to 12 months as clinically indicated. Adherence to both medication and lifestyle regimens are required for ASCVD risk reduction. After statin therapy has been initiated, some

<sup>†</sup>In those already on a statin, in whom baseline LDL-C is unknown, an LDL-C level <100 mg/dL was observed in most individuals receiving high-intensity statin therapy

<sup>‡</sup>Clinical ASCVD includes acute coronary syndromes, or a history of myocardial infarction, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack, or peripheral arterial disease presumed to be of atherosclerotic origin.

ACC indicates American College of Cardiology; AHA, American Heart Association; ASCVD, atherosclerotic cardiovascular disease; COR, Class of Recommendation; LDL-C, low-density lipoprotein cholesterol; LOE, Level of Evidence; NHLBI, National Heart, Lung, and Blood Institute; RCTs, randomized controlled trials; and —, not applicable.



Figure 5. Statin Therapy: Monitoring Therapeutic Response and Adherence

Colors correspond to the Classes of Recommendation in Table 1.

\*Fasting lipid panel preferred. In a nonfasting individual, a non–HDL-C level ≥220 mg/dL may indicate genetic hypercholesterolemia that requires further evaluation or a secondary etiology. If nonfasting triglycerides are ≥500 mg/dL, a fasting lipid panel is required.

†In those already on a statin, in whom baseline LDL-C is unknown, an LDL-C <100 mg/dL was observed in most individuals receiving high-intensity statin therapy in RCTs. ±See Section 6.3.1.

HDL-C indicates high-density lipoprotein cholesterol; LDL-C, low-density lipoprotein cholesterol; and RCTs, randomized clinical trials.

individuals experience unacceptable adverse effects when taking the recommended intensity of statin therapy. Once the severity and association of adverse effects with statin therapy has been established, and once factors potentially contributing to statin intolerance are resolved, the patient should be given lower doses of the same statin or an alternative appropriate statin, until a statin and dose that have no adverse effects have been identified (Table 8, Recommendation 8).

See Figure 5 for a flow diagram on monitoring statin response for the initiation of nonstatin therapy.

#### **6.2. Optimizing Statin Therapy**

Although high-intensity statin therapy reduces ASCVD events more than moderate-intensity statin therapy, lower-intensity statin therapy has also been shown to reduce ASCVD events, although to a lesser degree. Therefore, individuals who merit guideline-recommended statin therapy should be treated with the maximum-appropriate intensity of a statin that does not cause adverse effects.

#### 6.3. Insufficient Response to Statin Therapy

#### 6.3.1. Testing

The evidence is less clear with regard to the most appropriate tests for determining whether an anticipated therapeutic response to statin therapy has occurred on the maximally tolerated dose. RCT evidence to support the use of specific LDL-C or non–HDL-C targets was not identified. The focus is on the intensity of the statin therapy, but as an aid to monitoring response to therapy and adherence, it is reasonable to use the following as indicators of anticipated therapeutic response to statin therapy:

- High-intensity statin therapy generally results in an average LDL-C reduction of ≥50% from the untreated baseline.
- Moderate-intensity statin therapy generally results in an average LDL-C reduction of 30% to <50% from the untreated baseline.
- LDL-C levels and percent reduction are to be used only to assess response to therapy and adherence.
   They are not to be used as performance standards.

In those already on a statin, in whom the baseline LDL-C is unknown, an LDL-C <100 mg/dL was observed in most individuals receiving high-intensity statin therapy in RCTs.

However, there are many limitations of using LDL-C <100 mg/dL as a fixed target. If a moderate- or low-intensity statin results in an LDL-C level <100 mg/dL in a patient with ASCVD, the evidence suggests that a high-intensity statin, if tolerated, provides a greater reduction in ASCVD events. Conversely, in those with LDL-C levels slightly >100 mg/dL on a high-intensity statin, some options such as niacin might require down-titration of the statin intensity in an effort to improve safety. This would result in a suboptimal intensity of evidence-based statin therapy. Additional limitations to using LDL-C treatment targets are discussed in the Full Panel Report Supplement.

No evidence was found that titration or combination-drug therapy to achieve specific LDL-C or non-HDL-C levels or percent reductions improved ASCVD outcomes. Therefore, this guideline does not recommend their use as performance measures.

The percent LDL-C reduction may not only indicate adherence, but also may reflect biological variability in the response to statin therapy. This acknowledges that some individuals may have less than an average response. Attention to adherence of statin and lifestyle therapy and evaluation and treatment of secondary causes (Table 6) that might elevate LDL-C, may address less-than-anticipated responses to a specific statin dosage. Whether the dose of statin therapy should be increased on the basis of a less-than-anticipated average response should be left to clinical judgment.

### 6.3.2. Nonstatins Added to Statins or in Statin-Intolerant Individuals

Adherence to lifestyle changes and to statin therapy should be reemphasized before the addition of a nonstatin drug is considered (Figure 5). RCTs evaluating the ASCVD event reductions from nonstatins used as monotherapy were reviewed, as were RCTs evaluating the additional reduction in ASCVD events from nonstatin therapy added to statin therapy. The Expert Panel could find no data supporting the routine use of nonstatin drugs combined with statin therapy to further reduce ASCVD events. In addition, no RCTs that assessed ASCVD outcomes in statin-intolerant patients were found.

Clinicians treating high-risk patients who have a less-than-anticipated response to statins, who are unable to tolerate a less-than-recommended intensity of a statin, or who are completely statin intolerant, may consider the addition of a nonstatin cholesterol-lowering therapy. High-risk individuals include those with ASCVD, those with LDL-C ≥190 mg/dL, and those with diabetes 40–75 years of age. In this situation, this guideline recommends clinicians preferentially prescribe drugs that have been shown in RCTs to provide ASCVD risk-reduction benefits that outweigh the potential for adverse

effects and drug-drug interactions, and consider patient preferences.

### 7. Selected Clinical and Population Subgroups

#### 7.1. Sex and Racial and Ethnic Subgroups

Because the RCT evidence shows that the absolute benefit of statin treatment is proportional to baseline ASCVD risk, treatment decisions for women and racial and ethnic subgroups should be based on the level of ASCVD risk. This conclusion is a departure from previous approaches that focused on LDL-C levels to guide treatment decisions. Statin treatment based on estimated 10-year ASCVD risk avoids the overtreatment of lower-risk groups, such as younger, non-Hispanic white women who, despite moderate elevations in LDL-C, are typically not at significantly increased risk for ASCVD in the next 10 years in the absence of substantial risk factor burden. However, ignoring the increased ASCVD risk in African American women and men might result in the undertreatment of some individuals who are at significantly higher ASCVD risk at the same LDL-C level. Thus, this guideline recommends statin therapy for individuals in whom it is most likely to provide ASCVD risk reduction on the basis of the estimated 10-year risk of ASCVD.

#### 7.2. Individuals >75 Years of Age

Fewer people >75 years of age were enrolled in the statin RCTs reviewed. RCT evidence does support the continuation of statins beyond 75 years of age in persons who are already taking and tolerating these drugs. A larger amount of data supports the use of moderate-intensity statin therapy for secondary prevention in individuals with clinical ASCVD who are >75 years of age. However, the limited information available did not clearly support initiation of high-intensity statin therapy for secondary prevention in individuals >75 years of age.

Few data were available to indicate an ASCVD event reduction benefit in primary prevention among individuals >75 years of age who do not have clinical ASCVD. Therefore, initiation of statins for primary prevention of ASCVD in individuals >75 years of age requires consideration of additional factors, including increasing comorbidities, safety considerations, and priorities of care. The Pooled Cohort Equations can also provide information on expected 10-year ASCVD risk for those 76 to 79 years of age that may inform the treatment decision. These factors may influence decisions about cholesterol-lowering drug therapy, especially in the primary-prevention setting. Accordingly, a discussion of the potential ASCVD riskreduction benefits, risk of adverse effects, drug-drug interactions, and consideration of patient preferences should precede the initiation of statin therapy for primary prevention in older individuals.

#### 8. Limitations

The evidence-based recommendations in this guideline focus on patient groups who are well represented in RCTs and/or are highly likely to have high-risk genetic conditions, so the recommendations are designed to inform rather than replace clinical judgment. However, there are other patient groups for which a robust evidence base is lacking but that may nevertheless include some persons for whom statin treatment should be considered (after taking patient preferences into account) on the basis of the potential for ASCVD benefits to exceed the risk of adverse events and drug-drug interactions. Clinician judgment is especially important for several patient groups for which the RCT evidence is insufficient for guiding clinical recommendations. These patient groups include younger adults (<40 years of age) who have a low estimated 10-year ASCVD risk but a high lifetime ASCVD risk based on single strong factors or multiple risk factors. Other groups include those with serious comorbidities and increased ASCVD risk (e.g., individuals with HIV or rheumatologic or inflammatory diseases, or who have undergone a solid organ transplantation). This guideline encourages clinicians to use clinical judgment in these situations, weighing potential benefits, adverse effects, drug-drug interactions, and consider patient preferences.

Previous guidelines have taken less rigorous approaches to identifying the evidence to support their recommendations. In contrast, to minimize various sources of bias, the present recommendations are based on data available from RCTs and systematic reviews and meta-analyses of RCTs that were graded as fair to good quality by an independent contractor and were reviewed by the Expert Panel, with the assistance of an independent methodologist. To avoid biases, evidence from post-hoc analyses of included RCTs, from poor-quality RCTs, and from observational studies was not considered. This approach resulted in a comprehensive set of evidence-based clinical recommendations for the treatment of blood cholesterol to reduce ASCVD risk.

### 9. Evidence Gaps and Future Research Needs

After a systematic review of the literature, several research priorities are suggested that address existing evidence gaps and offer the greatest potential to inform and influence clinical practice and reduce ASCVD morbidity and mortality. High-priority research areas are:

- 1. Outcomes of RCTs to evaluate statins for the primary prevention of ASCVD in adults >75 years of age.
- 2. Outcomes of RCTs to evaluate alternative treatment strategies for ASCVD risk reduction. These RCTs

- may compare titration to specific cholesterol or apolipoprotein goals versus fixed-dose statin therapy in high-risk patients.
- RCTs to determine whether submaximal statin doses, combined with nonstatin therapies, reduce ASCVD risk in statin-intolerant patients.
- 4. Evaluation of the incidence, pathophysiology, clinical course, and clinical outcomes of new-onset diabetes associated with statin therapy.
- Outcomes of RCTs of new lipid-modifying agents to determine the incremental ASCVD event-reduction benefits when added to evidence-based statin therapy.

Additional research recommendations are included in the Full Panel Report Supplement.

#### 10. Conclusions

These recommendations arose from careful consideration of an extensive body of higher-quality evidence derived from RCTs and systematic reviews and meta-analyses of RCTs. Rather than LDL-C or non-HDL-C targets, this guideline used the intensity of statin therapy as the goal of treatment. Through a rigorous process, 4 groups of individuals were identified for whom an extensive body of RCT evidence demonstrated a reduction in ASCVD events with a good margin of safety from moderate- or high-intensity statin therapy:

#### Four Statin Benefit Groups:

- 1. Individuals with clinical ASCVD
- 2. Individuals with primary elevations of LDL-C  $\geq$ 190 mg/dL
- 3. Individuals 40 to 75 years of age with diabetes and LDL-C 70 to 189 mg/dL without clinical ASCVD
- 4. Individuals without clinical ASCVD or diabetes who are 40 to 75 years of age and have LDL-C 70 to 189 mg/dL and an estimated 10-year ASCVD risk of ≥7.5%. This requires a clinician-patient discussion.

Individuals in the last group can be identified by using the Pooled Cohort Equations for ASCVD risk prediction developed by the Risk Assessment Work Group. Lifestyle counseling should occur at the initial and follow-up visits as the foundation for statin therapy and may improve the overall risk factor profile.

Most importantly, our focus is on those individuals most likely to benefit from evidence-based statin therapy to reduce ASCVD risk. Implementation of these ASCVD risk-reduction guidelines will help to substantially address the large burden of fatal and nonfatal ASCVD in the United States. We realize that these guidelines represent a change from previous guidelines, but clinicians have become accustomed to change when that change is consistent with the current evidence. Continued accumulation of quality trial data will inform future cholesterol treatment guidelines.
#### **Presidents and Staff**

#### American College of Cardiology

John Gordon Harold, MD, MACC, President Shalom Jacobovitz, Chief Executive Officer William J. Oetgen, MD, MBA, FACC, Executive Vice President, Science, Education, & Quality Charlene May, Senior Director, Science and Clinical Policy

American College of Cardiology/American Heart Association Lisa Bradfield, CAE, Director, Science and Clinical Policy Emily Schiller, Specialist, Science and Clinical Policy

#### American Heart Association

Mariell Jessup, MD, FACC, FAHA, President Nancy Brown, Chief Executive Officer Rose Marie Robertson, MD, FAHA, Chief Science

Gayle R. Whitman, PhD, RN, FAHA, FAAN, Senior Vice President, Office of Science Operations

Marco Di Buono, PhD, Vice President of Science and Research

Jody Hundley, Production Manager, Scientific Publications, Office of Science Operations

National Heart, Lung, and Blood Institute Glen Bennett, MPH Denise Simons-Morton, MD, PhD

#### REFERENCES

- Institute of Medicine (U.S.) Committee on Standards for Developing Trustworthy Clinical Practice Guidelines, Graham R. Clinical Practice Guidelines We Can Trust. Washington, D.C.: National Academies Press; 2011.
- Gibbons GH, Harold JG, Jessup M, et al. The next steps in developing clinical practice guidelines for prevention. J Am Coll Cardiol 2013;62:1399–400.
- 3. Gibbons GH, Shurin SB, Mensah GA, et al. Refocusing the agenda on cardiovascular guidelines: an announcement from the National Heart, Lung, and Blood Institute. Circulation 2013;128: 1713-5
- Expert Panel on Integrated Guidelines for Cardiovascular Health and Risk Reduction in Children and Adolescents, National Heart Lung and Blood Institute. Expert panel on integrated guidelines for cardiovascular health and risk reduction in children and adolescents: summary report. Pediatrics 2011;128 Suppl 5:S213–56.
- Yancy CW, Jessup M, Bozkurt B, et al. 2013 ACCF/AHA guideline for the management of heart failure: executive summery: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol 2013;62:1495–539.
- National Cholesterol Education Program (U.S.), National Heart, Lung, and Blood Institute, National Institutes of Health. Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) Final Report. Bethesda, MD: National Cholesterol Education Program, National Heart, Lung, and Blood Institute, National Institutes of Health; 2002. NIH Publication No. 02–5215.
- Grundy S, Cleeman J, Merz C, et al. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III guidelines. Circulation 2004;110:227–39.
- 8. National Cholesterol Education Program (U.S.) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in

- Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adults Treatment Panel III) Final report. Circulation 2002; 106:3143–421.
- AIM-HIGH Investigators, Boden WE, Probstfield JL. Niacin in patients with low HDL cholesterol levels receiving intensive statin therapy. N Engl J Med 2011;67:2255–67.
- Eckel RH, Jakicic JM, Ard JD, et al. 2013 AHA/ACC guideline on lifestyle management to reduce cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol 2014;63: 2960–84.
- Goff DC Jr., Lloyd-Jones DM, D'Agostino RB Sr., et al. 2013 ACC/AHA guideline on the assessment of cardiovascular risk. J Am Coll Cardiol 2014;63:2935–59.
- Taylor F, Huffman MD, Macedo AF, et al. Statins for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev 2013.
- Cholesterol Treatment Trialists' (CTT) Collaborators, Mihaylova B, Emberson J, et al. The effects of lowering LDL cholesterol with statin therapy in people at low risk of vascular disease: meta-analysis of individual data from 27 randomised trials. Lancet 2012;380: 581–90.
- ACCORD Study Group, Ginsberg HN, Elam MB, et al. Effects of combination lipid therapy in type 2 diabetes mellitus. N Engl J Med 2010;362:1563–74.
- Taylor F, Ward K, Moore TH, et al. Statins for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev 2011. CD004816.
- Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. Lancet 2002;360:7–22.
- Downs JR, Clearfield M, Weis S, et al. Primary prevention of acute coronary events with lovastatin in men and women with average cholesterol levels: results of AFCAPS/TexCAPS. Air Force/ Texas Coronary Atherosclerosis Prevention Study. JAMA 1998; 279:1615–22.
- Nakamura H, Arakawa K, Itakura H, et al. Primary prevention of cardiovascular disease with pravastatin in Japan (MEGA Study): a prospective randomised controlled trial. Lancet 2006;368: 1155–63.
- Lu Z, Kou W, Du B, et al. Effect of Xuezhikang, an extract from red yeast Chinese rice, on coronary events in a Chinese population with previous myocardial infarction. Am J Cardiol 2008;101: 1689–93.
- Cholesterol Treatment Trialists' (CTT) Collaboration, Baigent C, Blackwell L. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet 2010;376:1670–81.
- 21. Tikkanen MJ, Holme I, Cater NB, et al. Comparison of efficacy and safety of atorvastatin (80 mg) to simvastatin (20 to 40 mg) in patients aged <65 versus >or=65 years with coronary heart disease (from the Incremental Decrease through Aggressive Lipid Lowering [IDEAL] study). Am J Cardiol 2009;103:577–82.
- Holmes HM, Hayley DC, Alexander GC, et al. Reconsidering medication appropriateness for patients late in life. Arch Intern Med 2006;166:605–9.
- Akushevich I, Kravchenko J, Ukraintseva S, et al. Age patterns of incidence of geriatric disease in the U.S. elderly population: Medicare-based analysis. J Am Geriatr Soc 2012;60:323–7.
- Wolff JL, Starfield B, Anderson G. Prevalence, expenditures, and complications of multiple chronic conditions in the elderly. Arch Intern Med 2002;162:2269–76.
- Fried TR, Tinetti ME, Towle V, et al. Effects of benefits and harms on older persons' willingness to take medication for primary cardiovascular prevention. Arch Intern Med 2011;171:923–8.
- Robinson JG, Bakris G, Torner J, et al. Is it time for a cardiovascular primary prevention trial in the elderly? Stroke 2007;38:441–50.
- Porock D, Oliver D, Zweig S, et al. Predicting death in the nursing home: development and validation of the 6-month Minimum Data Set mortality risk index. J Gerontol A Biol Sci Med Sci 2005;60: 491–8.

Stone et al.

- Stineman MG, Xie D, Pan Q, et al. All-cause 1-, 5-, and 10-year mortality in elderly people according to activities of daily living stage. J Am Geriatr Soc 2012;60:485–92.
- Schonberg MA, Davis RB, McCarthy EP, et al. External validation of an index to predict up to 9-year mortality of community-dwelling adults aged 65 and older. J Am Geriatr Soc 2011;59:1444–51.
- Fried TR, Tinetti ME, Iannone L, et al. Health outcome prioritization as a tool for decision making among older persons with multiple chronic conditions. Arch Intern Med 2011;171:1854–6.
- 31. Barry MJ, Edgman-Levitan S. Shared decision making—pinnacle of patient-centered care. N Engl J Med 2012;366:780–1.
- Man-Son-Hing M, Gage B, Montgomery AA. Preference-based antithrombotic therapy in atrial fibrillation: implications for clinical decision making. Med Decis Making 2005;25:548–59.
- Fried TR, Bradley EH, Towle VR, et al. Understanding the treatment preferences of seriously ill patients. N Engl J Med 2002;346: 1061–6.
- 34. Ditto PH, Druley JA, Moore KA, et al. Fates worse than death: the role of valued life activities in health-state evaluations. Health Psychol 1996;15:332–43.
- 35. Rosenfeld KE, Wenger NS, Kagawa-Singer M. End-of-life decision making: a qualitative study of elderly individuals. J Gen Intern Med 2000;15:620–5.
- Nease RJ, Kneeland T, O'Connor GT, et al. Variation in patient utilities for outcomes of the management of chronic stable angina: Implications for clinical practice guidelines. Ischemic Heart Disease Patient Outcomes Research Team. JAMA 1995;273:1185–90.
- 37. Glynn RJ, Koenig W, Nordestgaard BG, et al. Rosuvastatin for primary prevention in older persons with elevated C-reactive protein and low to average low-density lipoprotein cholesterol levels: exploratory analysis of a randomized trial. Ann Int Med 2010;152: 488–96. W174.
- Shepherd J, Blauw GJ, Murphy MB, et al. Pravastatin in elderly individuals at risk of vascular disease (PROSPER): a randomised controlled trial. Lancet 2002;360:1623–30.
- Trompet S, van Vliet P, de Craen AJM, et al. Pravastatin and cognitive function in the elderly. Results of the PROSPER study. J Neurol 2010;257:85–90.
- Gray SL, Boudreau RM, Newman AB, et al. Angiotensinconverting enzyme inhibitor and statin use and incident mobility limitation in community-dwelling older adults: the Health, Aging and Body Composition Study. J Am Geriatr Soc 2011;59: 2226–32.
- 41. LaCroix AZ, Gray SL, Aragaki A, et al. Statin use and incident frailty in women aged 65 years or older: prospective findings from the Women's Health Initiative Observational Study. J Gerontol A Biol Sci Med Sci 2008;63:369–75.
- Hippisley-Cox J, Pringle M, Cater R, et al. Coronary heart disease prevention and age inequalities: the first year of the National Service Framework for CHD. Br J Gen Pract 2005;55:369–75.
- Forman DE, Rich MW, Alexander KP, et al. Cardiac care for older adults. Time for a new paradigm. J Am Coll Cardiol 2011;57: 1801–10.
- Berglund L, Brunzell JD, Goldberg AC, et al. Evaluation and treatment of hypertriglyceridemia: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab 2012;97:2969–89.
- Miller M, Stone NJ, Ballantyne C, et al. Triglycerides and cardiovascular disease: a scientific statement from the American Heart Association. Circulation 2011;123:2292–333.
- LaRosa JC, Grundy SM, Waters DD, et al. Intensive lipid lowering with atorvastatin in patients with stable coronary disease. N Engl J Med 2005;352:1425–35.
- Pedersen TR, Faergeman O, Kastelein JJP, et al. High-dose atorvastatin vs usual-dose simvastatin for secondary prevention after myocardial infarction: the IDEAL study: a randomized controlled trial. JAMA 2005;294:2437–45.
- Cannon CP, Braunwald E, McCabe CH, et al. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med 2004;350:1495–504.
- Ridker PM, Danielson E, Fonseca FAH, et al. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med 2008;359:2195–207.
- 50. Baigent C, Keech A, Kearney P, et al. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data

- from 90,056 participants in 14 randomised trials of statins. Lancet 2005;366:1267–78.
- 51. Thompson GR, Packard CJ, Stone NJ. Goals of statin therapy: three viewpoints. 2002. Atheroscler Suppl 2004;5:107–14.
- Ridker PM, Pradhan A, MacFadyen JG, et al. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet 2012;380:565–71.
- Roffi M, Angiolillo DJ, Kappetein AP. Current concepts on coronary revascularization in diabetic patients. Eur Heart J 2011;32: 2748–57.
- Nathan DM, Cleary PA, Backlund JY, et al. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med 2005;353:2643–53.
- Rhodes ET, Prosser LA, Hoerger TJ, et al. Estimated morbidity and mortality in adolescents and young adults diagnosed with Type 2 diabetes mellitus. Diabet Med 2012;29:453–63.
- Paynter NP, Mazer NA, Pradhan AD, et al. Cardiovascular risk prediction in diabetic men and women using hemoglobin A1c vs diabetes as a high-risk equivalent. Arch Intern Med 2011;171:1712–8.
- 57. Elley CR, Robinson E, Kenealy T, et al. Derivation and validation of a new cardiovascular risk score for people with type 2 diabetes: the New Zealand Diabetes Cohort Study. Diabetes Care 2010;33: 1347–52.
- Stevens RJ, Coleman RL, Adler AI, et al. Risk factors for myocardial infarction case fatality and stroke case fatality in type 2 diabetes: UKPDS 66. Diabetes Care 2004;27:201–7.
- Bibbins-Domingo K, Coxson P, Pletcher MJ, et al. Adolescent overweight and future adult coronary heart disease. N Engl J Med 2007;357:2371–9.
- Daniels SR, Jacobson MS, McCrindle BW, et al. American Heart Association Childhood Obesity Research Summit Report. Circulation 2009;119:e489–517.
- Jacob M, Cho L. Asian Americans and cardiometabolic risk: why and how to study them. J Am Coll Cardiol 2010;55:974–5.
- Bainey KR, Jugdutt BI. Increased burden of coronary artery disease in South-Asians living in North America. Need for an aggressive management algorithm. Atherosclerosis 2009;204:1–10.
- 63. Yu T, Vollenweider D, Varadhan R, et al. Support of personalized medicine through risk-stratified treatment recommendations an environmental scan of clinical practice guidelines. BMC Med 2013; 11.7
- Lescol (fluvastatin sodium) [prescribing information]. Novartis Pharmaceuticals. East Hanover, NJ; 2012.
- 65. Pravachol (pravastatin sodium) [prescribing information]. Bristol Myers Squibb Co. Princeton, NJ; 2012.
- Livalo (pitivastatin) [prescribing information]. Kowa Pharmaceuticals. Montgomery, AL; 2012.
- 67. Zocor (Simvastatin) [prescribing information]. Merck & Co. Whitehouse Station, NJ; 2012.
- 68. Mevacor (Lovastatin) [prescribing information]. Merck & Co. Whitehouse Station, NJ; 2012.
- Lipitor (atorvastatin calcium) [prescribing information]. Pfizer Inc. New York, NY; 2012.
- Crestor (rosuvastatin calcium) [prescribing information]. AstraZeneca Pharmaceuticals. Wilmington, DE; 2013.
- Randomised trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S). Lancet 1994;344:1383–9.
- Shepherd J, Cobbe SM, Ford I, et al. Prevention of coronary heart disease with pravastatin in men with hypercholesterolemia. West of Scotland Coronary Prevention Study Group. N Engl J Med 1995; 333:1301–7.
- Sacks FM, Pfeffer MA, Moye LA. The effect of pravastatin on coronary events after myocardial infarction in patients with average cholesterol levels. Cholesterol and Recurrent Events Trial investigators. N Engl J Med 1996;335:1001–9.
- 74. Prevention of cardiovascular events and death with pravastatin in patients with coronary heart disease and a broad range of initial cholesterol levels. The Long-Term Intervention with Pravastatin in Ischaemic Disease (LIPID) Study Group. N Engl J Med 1998;339: 1349–57.
- Colhoun HM, Betteridge DJ, Durrington PN, et al. Primary prevention of cardiovascular disease with atorvastatin in type 2 diabetes in the Collaborative Atorvastatin Diabetes Study (CARDS):

- multicentre randomised placebo-controlled trial. Lancet 2004;364: 685-96.
- 76. Deleted in Press.
- Amarenco P, Bogousslavsky J, Callahan Ar, et al. High-dose atorvastatin after stroke or transient ischemic attack. N Engl J Med 2006;355:549–59.
- The Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) Investigators. High-dose atorvastatin after stroke or transient ischemic attack. N Engl J Med 2006;355:549–59.
- Vodnala D, Rubenfire M, Brook RD. Secondary causes of dyslipidemia. Am J Cardiol 2012;110:823–5.
- Stone NJ, Blum CB. Management of Lipids in Clinical Practice. 7th ed. Caddo, OK: Professional Communications; 2008.
- 81. Sattar N, Preiss D, Murray HM, et al. Statins and risk of incident diabetes: a collaborative meta-analysis of randomised statin trials. Lancet 2010;375:735–42.
- 82. Guiding the guidelines. Lancet 2011;377:1125.
- 83. Expert Panel on Detection Evaluation and Treatment of High Blood Cholesterol in Adults. Executive Summary of the Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). JAMA 2001;285:2486–97.
- Fellström BC, Jardine AG, Schmieder RE, et al. Rosuvastatin and cardiovascular events in patients undergoing hemodialysis. N Engl J Med 2009;360:1395–407.
- 85. Kjekshus J, Apetrei E, Barrios V, et al. Rosuvastatin in older patients with systolic heart failure. N Engl J Med 2007;357:2248–61.
- Gissi-HF Investigators, Tavazzi L, Maggioni AP, et al. Effect of rosuvastatin in patients with chronic heart failure (the GISSI-HF trial): a randomised, double-blind, placebo-controlled trial. Lancet 2008;372:1231–9.
- 87. Wanner C, Krane V, März W, et al. Atorvastatin in patients with type 2 diabetes mellitus undergoing hemodialysis. N Engl J Med 2005;353:238–48.
- 88. Eckel RH. Approach to the patient who is intolerant of statin therapy. J Clin Endocrinol Metab 2010;95:2015–22.
- U.S. Food and Drug Administration. FDA Drug Safety Communication: important safety label changes to cholesterol-lowering statin drugs. Rockville, MD: U.S. Food and Drug Administration; 2012.
- U.S. Food and Drug Administration. FDA Drug Safety Communication: ongoing safety review of high-dose Zocor (simvastatin) and increased risk of muscle injury. Rockville, MD: U.S. Food and Drug Administration; 2010.
- Association AD. Standards of medical care in diabetes–2013. Diabetes Care 2013;36 Suppl 1:S11–66.
- 92. Rawlins M. De testimonio: on the evidence for decisions about the use of therapeutic interventions. Lancet 2008;372:2152–61.
- Schwartz GG, Olsson AG, Ezekowitz MD, et al. Effects of atorvastatin on early recurrent ischemic events in acute coronary syndromes: the MIRACL study: a randomized controlled trial. JAMA 2001;285:1711–8.
- 94. Shepherd J, Barter P, Carmena R, et al. Effect of lowering LDL cholesterol substantially below currently recommended levels in patients with coronary heart disease and diabetes: the Treating to New Targets (TNT) study. Diabetes Care 2006;29: 1220–6.
- 95. Deleted in Press.
- Baigent C, Blackwell L, Emberson J, et al. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet 2010;376: 1670–81.
- Mills EJ, Rachlis B, Wu P, et al. Primary prevention of cardiovascular mortality and events with statin treatments: a network metaanalysis involving more than 65,000 patients. J Am Coll Cardiol 2008;52:1769–81.
- Dale KM, White CM, Henyan NN, et al. Impact of statin dosing intensity on transaminase and creatine kinase. Am J Med 2007;120: 706–12.
- 99. Collins R, Armitage J, Parish S, et al. Effects of cholesterol-lowering with simvastatin on stroke and other major vascular events in 20536 people with cerebrovascular disease or other high-risk conditions. Lancet 2004;363:757–67.

- Roberts MD. Crestor (rosuvastatin calcium) NDA 21–336 JUPITER. Paper presented at U.S. Food and Drug Administration, Endocrinologic and Metabolic Drugs Advisory Meeting, December 15, 2009. Gaithersburg, MD: U.S. Food and Drug Administration; 2009.
- Clofibrate and niacin in coronary heart disease. JAMA 1975;231: 360–81.
- Guyton JR, Bays HE. Safety considerations with niacin therapy. Am J Cardiol 2007;99:22C–31C.
- Brown BG, Zhao XQ. Nicotinic acid, alone and in combinations, for reduction of cardiovascular risk. Am J Cardiol 2008; 101:58B-62B.
- 104. Grundy SM, Vega GL, McGovern ME, et al. Efficacy, safety, and tolerability of once-daily niacin for the treatment of dyslipidemia associated with type 2 diabetes: results of the assessment of diabetes control and evaluation of the efficacy of niaspan trial. Arch Intern Med 2002;162:1568–76.
- Crouse JR 3rd Hypertriglyceridemia: a contraindication to the use of bile acid binding resins. Am J Med 1987;83:243–8.
- Thompson GR, HEART-UK LDL Apheresis Working Group. Recommendations for the use of LDL apheresis. Atherosclerosis 2008;198:247–55.
- Schwertz DW, Badellino KO. High-dose statin therapy for secondary prevention of stroke: stroke prevention by aggressive reduction in cholesterol levels study review. J Cardiovasc Nurs 2008; 23:8–13.
- Rossebo AB, Pedersen TR, Allen C, et al. Design and baseline characteristics of the Simvastatin and Ezetimibe in Aortic Stenosis (SEAS) study. Am J Cardiol 2007;99:970–3.
- 109. Sharp Collaborative Group. Study of Heart and Renal Protection (SHARP): randomized trial to assess the effects of lowering lowdensity lipoprotein cholesterol among 9,438 patients with chronic kidney disease. Am Heart J 2010;160:785–794. e10.
- 110. Yokoyama M, Origasa H, JELIS Investigators. Effects of eicosapentaenoic acid on cardiovascular events in Japanese patients with hypercholesterolemia: rationale, design, and baseline characteristics of the Japan EPA Lipid Intervention Study (JELIS). Am Heart J 2003;146:613–20.
- 111. Frick MH, Elo O, Haapa K, et al. Helsinki Heart Study: primary-prevention trial with gemfibrozil in middle-aged men with dyslipidemia. Safety of treatment, changes in risk factors, and incidence of coronary heart disease. N Engl J Med 1987;317:1237–45.
- 112. The Lipid Research Clinics Coronary Primary Prevention Trial results. II. The relationship of reduction in incidence of coronary heart disease to cholesterol lowering. JAMA 1984;251:365–74.
- The Lipid Research Clinics Coronary Primary Prevention Trial results. I. Reduction in incidence of coronary heart disease. JAMA 1984;251:351–64.
- 114. Rubins HB, Robins SJ, Collins D, et al. Gemfibrozil for the secondary prevention of coronary heart disease in men with low levels of high-density lipoprotein cholesterol. Veterans Affairs High-Density Lipoprotein Cholesterol Intervention Trial Study Group. N Engl J Med 1999;341:410–8.
- 115. Keech A, Simes RJ, Barter P, et al. Effects of long-term fenofibrate therapy on cardiovascular events in 9795 people with type 2 diabetes mellitus (the FIELD study): randomised controlled trial. Lancet 2005;366:1849–61.
- 116. HPS2-THRIVE Collaborative Group. HPS2-THRIVE randomized placebo-controlled trial in 25 673 high-risk patients of ER niacin/laropiprant: trial design, pre-specified muscle and liver outcomes, and reasons for stopping study treatment. Eur Heart J 2013; 34:1279–91.
- 117. De Lemos JA, Blazing MA, Wiviott SD, et al. Early intensive vs a delayed conservative simvastatin strategy in patients with acute coronary syndromes: phase Z of the A to Z trial. JAMA 2004;292: 1307–16.
- 118. Koren MJ, Hunninghake DB, ALLIANCE Investigators. Clinical outcomes in managed-care patients with coronary heart disease treated aggressively in lipid-lowering disease management clinics: the ALLIANCE study. J Am Coll Cardiol 2004;44:1772–9.
- 119. Knopp RH, d' Emden M, Smilde JG, et al. Efficacy and safety of atorvastatin in the prevention of cardiovascular end points in subjects with type 2 diabetes: the Atorvastatin Study for Prevention of Coronary Heart Disease Endpoints in non-insulin-dependent diabetes mellitus (ASPEN). Diabetes Care 2006;29:1478–85.

Stone et al.

- 120. Athyros VG, Papageorgiou AA, Mercouris BR, et al. Treatment with atorvastatin to the National Cholesterol Educational Program goal versus "usual" care in secondary coronary heart disease prevention. The GREek Atorvastatin and Coronary-heart-disease Evaluation (GREACE) study. Curr Med Res Opin 2002;18:220–8.
- 121. Brown BG, Zhao XQ, Chait A, et al. Simvastatin and niacin, antioxidant vitamins, or the combination for the prevention of coronary disease. N Engl J Med 2001;345:1583–92.
- 122. Serruys PWJC, de Feyter P, Macaya C, et al. Fluvastatin for prevention of cardiac events following successful first percutaneous coronary intervention: a randomized controlled trial. JAMA 2002; 287:3215–22.
- 123. Sakamoto T, Kojima S, Ogawa H, et al. Effects of early statin treatment on symptomatic heart failure and ischemic events after acute myocardial infarction in Japanese. Am J Cardiol 2006;97: 1165–71.
- 124. Study of the Effectiveness of Additional Reductions in Cholesterol and Homocysteine (SEARCH) Collaborative Group, Armitage J, Bowman L, et al. Intensive lowering of LDL cholesterol with 80 mg versus 20 mg simvastatin daily in 12,064 survivors of myocardial infarction: a double-blind randomised trial. Lancet 2010; 376:1658–69.
- 125. Ahmed S, Cannon CP, Murphy SA, et al. Acute coronary syndromes and diabetes: is intensive lipid lowering beneficial? Results of the PROVE IT-TIMI 22 trial. Eur Heart J 2006;27:2323–9.
- 126. Wenger NK, Lewis SJ, Herrington DM, et al. Outcomes of using high- or low-dose atorvastatin in patients 65 years of age or older with stable coronary heart disease. Ann Int Med 2007;147: 1–9
- Chaturvedi S, Zivin J, Breazna A, et al. Effect of atorvastatin in elderly patients with a recent stroke or transient ischemic attack. Neurology 2009;72:688–94.
- 128. Shepherd J, Kastelein JJP, Bittner V, et al. Intensive lipid lowering with atorvastatin in patients with coronary heart disease and chronic kidney disease: The TNT (Treating to New Targets) study. J Am Coll Cardiol 2008;51:1448–54.
- 129. Shepherd J, Kastelein JP, Bittner VA, et al. Intensive lipid lowering with atorvastatin in patients with coronary artery disease, diabetes, and chronic kidney disease. Mayo Clin Proc 2008;83:870–9.
- 130. Sacks FM, Pfeffer MA, Moye LA, et al. The effect of pravastatin on coronary events after myocardial infarction in patients with average cholesterol levels. Cholesterol and Recurrent Events Trial Investigators. N Engl J Med 1996;335:1001–9.
- 131. ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. Major outcomes in moderately hypercholesterolemic, hypertensive patients randomized to pravastatin vs usual care: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT-LLT). JAMA 2002;288: 2998–3007.
- 132. Sever PS, Poulter NR, Dahlof B, et al. Reduction in cardiovascular events with atorvastatin in 2,532 patients with type 2 diabetes:

- Anglo-Scandinavian Cardiac Outcomes Trial-Lipid-Lowering Arm (ASCOT-LLA). Diabetes Care 2005;28:1151–7.
- 133. Holdaas H, Fellström B, Cole E, et al. Long-term cardiac outcomes in renal transplant recipients receiving fluvastatin: the ALERT extension study. Am J Transplant 2005;5:2929–36.
- 134. Cholesterol Treatment Trialists Collaboration, Kearney PM, Blackwell L, et al. Efficacy of cholesterol-lowering therapy in 18,686 people with diabetes in 14 randomised trials of statins: a metaanalysis. Lancet 2008;371:117–25.
- Messerli FH, Pinto L, Tang SSK, et al. Impact of systemic hypertension on the cardiovascular benefits of statin therapy—a metaanalysis. Am J Cardiol 2008;101:319–25.
- 136. Kizer JR, Madias C, Wilner B, et al. Relation of different measures of low-density lipoprotein cholesterol to risk of coronary artery disease and death in a meta-regression analysis of large-scale trials of statin therapy. Am J Cardiol 2010;105:1289–96.
- 137. Ray KK, Seshasai SRK, Erqou S, et al. Statins and all-cause mortality in high-risk primary prevention: a meta-analysis of 11 randomized controlled trials involving 65,229 participants. Arch Intern Med 2010;170:1024–31.
- 138. Brugts JJ, Yetgin T, Hoeks SE, et al. The benefits of statins in people without established cardiovascular disease but with cardiovascular risk factors: meta-analysis of randomised controlled trials. BMJ 2009;338:b2376.
- Bukkapatnam RN, Gabler NB, Lewis WR. Statins for primary prevention of cardiovascular mortality in women: a systematic review and meta-analysis. Prev Cardiol 2010;13:84–90.
- 140. Mizuno K, Nakaya N, Ohashi Y, et al. Usefulness of pravastatin in primary prevention of cardiovascular events in women: analysis of the Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese (MEGA study). Circulation 2008;117:494–502.
- 141. Bonovas S, Filioussi K, Tsantes A, et al. Use of statins and risk of haematological malignancies: a meta-analysis of six randomized clinical trials and eight observational studies. Br J Clin Pharmacol 2007;64:255–62.
- 142. Preiss D, Seshasai SRK, Welsh P, et al. Risk of incident diabetes with intensive-dose compared with moderate-dose statin therapy: a meta-analysis. JAMA 2011;305:2556-64.
- 143. Canner PL, Berge KG, Wenger NK, et al. Fifteen year mortality in Coronary Drug Project patients: long-term benefit with niacin. J Am Coll Cardiol 1986;8:1245–55.
- 144. Parolari A, Tremoli E, Cavallotti L, et al. Do statins improve outcomes and delay the progression of non-rheumatic calcific aortic stenosis? Heart 2011;97:523–9.

Key Words: ACC/AHA Practice Guideline ■ biomarkers, pharmacological ■ cardiovascular disease ■ cholesterol ■ diabetes mellitus ■ drug therapy ■ hydroxymethylglutaryl-CoA reductase inhibitors/statins ■ hypercholesterolemia ■ lipids ■ patient compliance ■ primary prevention ■ risk assessment ■ risk reduction behavior ■ secondary prevention.

# Appendix 1. Author Relationships With Industry and Other Entities (Relevant)—2013 ACC/AHA Guideline on the Treatment of Blood Cholesterol in Adults to Reduce Atherosclerotic Cardiovascular Risk

| Panel Member | Employment | Consultant | Speakers<br>Bureau | Ownership/<br>Partnership/<br>Principal | Personal<br>Research | Expert Witness |
|---|---|---|---|---|---|---|
| Neil J. Stone<br>Chair | Northwestern Memorial Hospital—Bonow Professor of Medicine, Feinberg School of Medicine, Northwestern University | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None |
| Jennifer G. Robinson<br>Co-Chair | University of lowa— Professor of Epidemiology and Medicine; Prevention Intervention Center—Director | 2008–2012:<br>None | 2008–2012:<br>None | <b>2008–2012:</b><br>None | 2008–2012: • Aegerion • Amarin* • Amgen* • AstraZeneca* • Esperion • Genentech/ Hoffman LaRoche* • GlaxoSmithKline* • Merck* • Sanofi-aventis/ Regeneron * | <b>2008–2012:</b><br>None |
| | | <b>2013:</b> None | <b>2013:</b><br>None | <b>2013</b> :<br>None | 2013: Amarin* Amgen* AstraZeneca* Genentech/ Hoffman LaRoche* GlaxoSmithKline* Merck* Sanofi-aventis/ Regeneron* | <b>2013:</b><br>None |
| Alice H. Lichtenstein<br>Co-Chair | Tufts University, USDA Human Nutrition Research Center on Aging—Gershoff Professor of Nutrition Science and Policy; Professor of Public Health and Family Medicine | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None |
| C. Noel Bairey Merz | Cedars-Sinai Medical Center—Women's Guild Endowed Chair in Women's Health Barbara Streisand Women's Heart Center—Director; Preventive Cardiac Center—Professor of Medicine | 2008–2012: • Abbott Vascular • Bayer • Bristol-Myers Squibb • Gilead • Novartis • Pfizer • Posen | 2008–2012:<br>None | 2008–2012: ATS Medical Boston Scientific Eli Lilly Johnson & Johnson Medtronic Teva Pharmaceuticals | 2008–2012: RWISE Ranexa Microvascular Ranexa Angina | <b>2008–2012:</b><br>None |
| | | 2013: • Amgen* • Gilead • Bristol-MyersSquibb (DSMB) | <b>2013:</b><br>None | <b>2013:</b><br>None | 2013:<br>• RWISE | <b>2013:</b><br>None |
| Conrad Blum | Columbia University Medical Center, Columbia University College of Physicians and Surgeons— Professor of Medicine | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None |

| Daniel Manahan | F1 | Oswanikant | Speakers | Ownership/<br>Partnership/ | Personal | F |
|---|---|---|---|---|---|---|
| Panel Member | Employment | Consultant | Bureau | Principal | Research | Expert Witness |
| Robert H. Eckel | University of Colorado, Denver School of Medicine—Professor of Medicine; Professor of Physiology and Biophysics; and Charles | 2008–2012: • Foodminds • Merck • Pfizer • Abbott | <b>2008–2012:</b><br>None | 2008–2012:<br>None | <b>2008–2012:</b><br>None | 2008–2012:<br>None |
| | A. Boettcher II Chair in<br>Atherosclerosis | 2013: • Amylin • Eli Lilly • Esperion • Foodminds • Johnson & Johnson • Novo Nordisk • Vivus | <b>2013:</b><br>None | <b>2013:</b><br>None | <ul><li>2013:</li><li>GlaxoSmithKline*</li><li>Sanofi-aventis/<br/>Regeneron</li></ul> | <b>2013:</b><br>None |
| Anne Carol Goldberg | Washington University<br>School of Medicine—<br>Associate Professor of<br>Medicine | 2008–2012: Abbott Roche ISIS/Genzyme Sanofi-aventis Unilever Merck | 2008–2012:<br>None | <b>2008–2012:</b><br>None | 2008-2012: Abbott* Aegerion* Amarin* Amgen* Genentech/Roche* GlaxoSmithKline* ISIS/Genzyme* Merck* Novartis Reliant* Sanofi-aventis/Regeneron* Sanofi-aventis* | 2008-2012:<br>None |
| | | 2013: • Merck | <b>2013:</b><br>None | <b>2013:</b><br>None | 2013: Abbott* Amarin* Amgen* Genentech/Roche* GlaxoSmithKline* ISIS/Genzyme* Merck* Sanofi-aventis/Regeneron* | 2013:<br>None |
| David Gordon, | NHLBI—Special Assistant | 2008–2012: | 2008–2012: | 2008-2012: | 2008–2012: | 2008-2012: |
| Ex-Officio | for Clinical Studies, | None | None | None | None | None |
| | Division of<br>Cardiovascular<br>Diseases | <b>2013:</b><br>None | <b>2013:</b><br>None | <b>2013:</b><br>None | <b>2013:</b><br>None | <b>2013:</b><br>None |
| Daniel Levy,<br>Ex-Officio | NHLBI—Director of the<br>Center for Population<br>Studies | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008-2012:<br>None<br>2013:<br>None |
| Donald M. Lloyd-Jones | Northwestern University<br>Feinberg School of<br>Medicine—Senior<br>Associate Dean; Chair<br>and Professor of<br>Preventive Medicine;<br>Professor of Medicine<br>(Cardiology) | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None |
| Patrick McBride | University of Wisconsin<br>School of Medicine and<br>Public Health—<br>Professor of Medicine<br>and Family Medicine | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None |

| Panel Member | Employment | Consultant | Speakers<br>Bureau | Ownership/<br>Partnership/<br>Principal | Personal<br>Research | Expert Witness |
|---|---|---|---|---|---|---|
| J. Sanford Schwartz | University of Pennsylvania<br>School of Medicine—<br>Leon Hess Professor of<br>Internal Medicine,<br>Health Management<br>and Economics | 2008–2012: Abbott Allergan Amgen Daiichi-Sankyo Genentech Johnson & Johnson Merck Pfizer Shire Pharmaceuticals | 2008–2012:<br>None | <b>2008–2012:</b><br>None | 2008–2012: • Pfizer | <b>2008–2012</b> :<br>None |
| | | 2013: Abbott Allergan Amgen Daiichi-Sankyo Genentech Johnson & Johnson Merck Pfizer Shire Pharmaceuticals | <b>2013:</b> None | <b>2013:</b><br>None | 2013: • Pfizer | <b>2013:</b><br>None |
| Susan T. Shero<br>Ex-Officio | NHLBI—Public Health<br>Advisor | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None |
| Sidney C. Smith, Jr | University of North Carolina—Professor of Medicine; Center for Cardiovascular Science and Medicine—Director | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None | 2008–2012:<br>None<br>2013:<br>None |
| Karol Watson | University of California,<br>Los Angeles School of<br>Medicine—Co-Director | 2008–2012: Abbott AstraZeneca Genzyme GlaxoSmithKline Kos Medtronic Merck Novartis Pfizer 2013: | 2008–2012:<br>None | 2008–2012:<br>None | 2008–2012: • Merck 2013: | 2008–2012:<br>None |
| | | 2013:<br>None | None | None | 2013:<br>● Merck | 2013:<br>None |
| Peter W.F. Wilson | Atlanta VA Medical Center | 2008–2012: | 2008–2012: | 2008–2012: | 2008–2012: | 2008–2012: |
| | and Emory University | Merck | None | None | Merck | None |
| | School of Medicine— | • XZK | | | <ul> <li>Liposcience</li> </ul> | |
| | Professor of Medicine | 2013: | 2013: | 2013: | 2013: | 2013: |
| | | None | None | None | <ul> <li>Merck</li> </ul> | None |

This table reflects the relevant healthcare-related relationships of authors with industry and other entities provided by the panels during the document development process (2008–2012). Both compensated and uncompensated relationships are reported. These relationships were reviewed and updated in conjunction with all meetings and conference calls of the Expert Panel during the document development process. Authors with relevant relationships during the document development process recused themselves from voting on recommendations relevant to their relationships. In the spirit of full transparency, the ACC and AHA asked Expert Panel members to provide updates and approve the final version of this table, which includes current relevant relationships (2013). To review the NHLBI and ACC/AHA's current comprehensive policies for managing relationships with industry and other entities, please refer to http://www.nhlbi.nih.gov/guidelines/cvd\_adult/coi-nvi\_policy.thm and http://www.cardiosource.org/Science-And-Quality/Practice-Guidelines-and-Quality-Standards/Relationships-With-Industry-Policy.aspx.  $Per\ ACC/AHA\ policy$ : A person is deemed to have a significant interest in a business if the interest represents ownership of  $\geq$ 5% of the voting stock or share of the business entity, or ownership of  $\geq$ 510,000 of the fair market value of the business entity; or if funds received by the person from the business entity exceed 5% of the person's gross income for the previous year. Relationships that exist with no financial benefit are also included for the purpose of transparency. Relationships in this table are modest unless otherwise noted.

 $* Significant\ relationship.\\$ 

ACC indicates American College of Cardiology; AHA, American Heart Association; NHLBI, National Heart, Lung, and Blood Institute; and USDA, U.S. Department of Agriculture.

# Appendix 2. Expert Reviewers Relationships With Industry and Other Entities—2013 ACC/AHA Guideline on the Treatment of Blood Cholesterol in Adults to Reduce Atherosclerotic Cardiovascular Risk

| Reviewer | Employment | Representation | Consultant | Speakers<br>Bureau | Ownership/<br>Partnership/<br>Principal | Personal<br>Research | Expert<br>Witness |
|---|---|---|---|---|---|---|---|
| Roger Blumenthal | Johns Hopkins Hospital Ciccarone Preventive Cardiology Center— Professor of Medicine | ACC/AHA | None | None | None | None | None |
| William Virgil Brown | Emory University School of Medicine | NLA | Abbott Amgen Anthera Bristol-Myers Squibb Catabasis Cerenis GlaxoSmithKline Genzyme LipoScience Merck Pfizer Regeneron | None | None | None | None |
| Linda Hemphill | Massachusetts General<br>Hospital—Director,<br>LDL Apheresis Program | NLA | Regeneron | None | None | None | None |
| Matthew Ito | Oregon Health & Science<br>University, Department<br>of Pharmacy Practice—<br>Professor | NLA | <ul><li>Aegeron</li><li>Kowa</li></ul> | None | None | None | None |
| Terry Jacobson | Emory University | NLA | <ul><li>Abbott</li><li>Merck</li></ul> | None | None | <ul><li>Amarin</li><li>HealthCore</li></ul> | None |
| Andrew Kates | Washington University School<br>of Medicine in St. Louis—<br>Cardiovascular Fellowship<br>Program Director | ACC/AHA | None | None | None | None | None |
| James M. McKenney | Virginia Commonwealth<br>University—Professor<br>Emeritus | NLA | None | None | None | None | None |
| E. Magnus Ohman | Duke Clinical Research<br>Institute—Professor of<br>Medicine; Program for<br>Advanced Coronary<br>Disease—Director | ACC/AHA Task<br>Force on<br>Practice<br>Guidelines | None | None | None | None | None |
| Carl E. Orringer | Case Western Reserve University<br>School of Medicine—Associate<br>Professor of Medicine | NLA | None | None | None | None | None |
| Robert S. Rosenson | Mount Sinai Hospital— Director, Preventive Cardiology; Professor of Medicine, Cardiology | NLA | <ul> <li>Amgen</li> <li>LipoScience</li> <li>Novartis</li> <li>Pfizer</li> <li>Sanofi-aventis/<br/>Regeneron</li> </ul> | None | • LipoScience | None | None |
| John Rumsfeld | Denver VA Medical Center, University of Colorado— National Director of Cardiology, U.S. Veterans Health Administration | ACC/AHA | None | None | None | None | None |
| Robert A. Wild | University of Oklahoma, College<br>of Medicine, Department of<br>Obstetrics and Gynecology—<br>Professor | NLA | Atherotec | None | None | None | None |

This table represents the relationships of reviewers with industry and other entities that were self-disclosed at the time of peer review. It does not necessarily reflect relationships with industry at the time of publication. To review the NHLBI and ACC/AHA's current comprehensive policies for managing relationships with industry and other entities, please refer to http://www.nhlbi.nih.gov/guidelines/cvd\_adult/coi-rwi\_policy.htm and http://www.cardiosource.org/Science-And-Quality/Practice-Guidelines-and-Quality-Standards/Relationships-With-Industry-Policy.aspx.

ACC indicates American College of Cardiology; AHA, American Heart Association; NLA, National Lipid Association; and VA, Veterans Affairs.

2923

## **Appendix 3. Abbreviations**

 $ALT = alanine \ transaminase$ 

 ${\sf ASCVD} = {\sf atherosclerotic\ cardiovascular\ disease}$ 

 $CHD = coronary\ heart\ disease$ 

COR = Class of Recommendation

 $\mathbf{CQ} = \mathbf{critical} \ \mathbf{question}$ 

 $\label{eq:hdl-constraint} \textbf{HDL-C} = \textbf{high-density lipoprotein cholesterol}$ 

 ${\bf LDL\text{-}C} = {\bf low\text{-}density} \ {\bf lipoprotein} \ {\bf cholesterol}$ 

LOE = Level of Evidence

 $\mathbf{MI} = \mathbf{myocardial}$  infarction

 ${\it NHLBI} = {\it National Heart, Lung, and Blood Institute}$ 

 $\label{eq:reconstruction} \textbf{RCT} = \textbf{randomized controlled trial}$ 

 $\label{eq:RWI} \textbf{RWI} = \textbf{relationships} \ \textbf{with} \ \textbf{industry} \ \textbf{and} \ \textbf{other} \ \textbf{entities}$ 

## **Appendix 4. Evidence Statements**

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 1 | Data are not available regarding treatment or titration to a specific LDL-C goal in adults with CHD/CVD. The Expert Panel found insufficient evidence to support setting LDL-C goals in CHD/CVD patients. | I | Secondary Prevention | Conclusion after reviewing 19 RCTs in CQ1 Evidence<br>Table:<br>4D (87), A-Z (117), ACCORD (14), ALLIANCE (118),<br>ASPEN (119), AURORA (84), CARE (73),<br>CORONA (85), GREACE (120), HATS (121), HPS<br>(16), IDEAL (47), LIPID (74), LIPS (122), MIRACL<br>(93), MUSHASHLAMI (123), PROVE-IT (48),<br>SPARCL (78,107), TNT (46) |
| 2 | The Expert Panel did not identify any trials in adults with CHD/CVD reporting mean or median on-treatment non-HDL-C levels in adults with CHD/CVD. | | Secondary Prevention | N/A |
| 3 | LDL-C goals <130 mg/dL or <100 mg/dL in patients without CHD/CVD. Randomized trial data are not available regarding dose titration to achieve a specific LDL-C goal. | I | Primary Prevention | Conclusion after reviewing 6 RCTs included in CQ2:<br>AFCAPS (17), ASPEN (119), AURORA (84), CARDS<br>(75), JUPITER (49), MEGA (18) |
| 4 | There was insufficient evidence in women without CHD/CVD to evaluate the reduction in CVD risk with achieved LDL-C levels $<$ 130 mg/dL or $<$ 100 mg/dL. | I | Primary Prevention | N/A |
| 5 | The Expert Panel did not identify any trials in adults without CHD/CVD reporting on-treatment non-HDL-C levels in adults with CHD/CVD. | | Primary Prevention | N/A |
| 6 | In adults with CHD/CVD, fixed high-intensity statin treatment (atorvastatin 40–80 mg) that achieved a mean LDL-C 67–79 mg/dL reduced the RR for CHD/CVD events more than fixed lower-dose statin treatment that achieved a mean LDL-C 97–102 mg/dL. In these trials, the mean LDL-C levels achieved differed by 23–30 mg/dL, or 22%–32%, between the 2 groups. Simvastatin 80 mg did not decrease CVD events compared with simvastatin 20–40 mg. See Table 4 for definitions of high, moderate, and low intensity for statins. Higher intensity = atorvastatin 40–80 mg Moderate intensity = atorvastatin 10 mg, pravastatin 40 mg, or simvastatin 20–40 mg | н | Secondary Prevention | Benefit: TNT (46), IDEAL (47), PROVE-IT (48) Lower LDL-C reductions, no benefit: A-Z (117), ACCORD (14) No difference in LDL-C between groups: (SEARCH (124) not included in CQ1) |
| 7 | In adults with CHD/CVD who do not have Class II-IV heart failure, fixed high-intensity statin (atorvastatin 80 mg) or statin-niacin treatment that achieved a mean LDL-C 72-79 mg/dL reduced the RR for CHD/CVD events compared with placebo with a mean LDL-C 112-135 mg/dL. In these trials, the mean LDL-C levels were reduced by 45-57 mg/dL or by 45% (HATS [121]) to 53% (SPARCL [107]). | н | Secondary Prevention | SPARCL (107) HATS (121) MIRACL (93) CORONA (85)-no benefit |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 8 | In adults with CHD/CVD and diabetes, fixed high-intensity statin treatment (atorvastatin 80 mg) that achieved a mean LDL-C of 57-77 mg/dL reduced the RR for CHD/CVD events more than fixed lower-intensity statin treatment that achieved a mean LDL-C of 81-99 mg/dL. In these trials, the mean LDL-C levels achieved differed by 22-24 mg/dL, or 22%-30%, between the 2 groups. | M to H | Secondary Prevention<br>(diabetes subgroup<br>included) | TNT (46,94), PROVE-IT (48,125)<br>No diabetes subgroup publications found for MIRACI<br>(93) or IDEAL (47) |
| 9 | In adults $\geq$ 65 years of age with CHD/CVD, fixed high-intensity statin treatment (atorvastatin 80 mg) that achieved a mean LDL-C of 72 mg/dL reduced CHD/CVD events more than fixed lower-intensity statin treatment that achieved a mean LDL-C of 97 mg/dL. In this trial, the mean LDL-C levels achieved differed by 25 mg/dL, or 26%, between the 2 groups. In adults $\geq$ 65 years of age with a history of stroke or TIA, higher fixed-dose statin treatment that achieved a mean LDL-C of 72 mg/dL reduced CHD events more than placebo, with a mean LDL-C of 129 mg/dL. In this trial, the mean LDL-C level was reduced by 61 mg/dL, or 46%, from baseline in those $\geq$ 65 years of age. | L | Secondary Prevention (age subgroups included) | TNT (46,126), SPARCL (107,127) No publications by age included for: PROVE-IT (48) IDEAL (47) HATS (121) |
| 10 | In adults with CHD/CVD and CKD (excluding hemodialysis), fixed high-<br>intensity statin treatment (atorvastatin 80 mg) that achieved a mean<br>LDL-C of 79 mg/dL reduced CHD/CVD events more than fixed lower-<br>dose statin treatment that achieved a mean LDL-C of 99 mg/dL. In this<br>trial, the mean LDL-C levels achieved differed by 20 mg/dL, or 20%<br>between the 2 groups. | L | Secondary Prevention (CKD subgroup included) | TNT (46,128) TNT (46,129) No publications included for CKD: PROVE-IT (48) IDEAL (47) |
| 11 | In adults with CHD or acute coronary syndromes, more intensive-dose statin therapy reduced LDL-C to a greater degree (by 20 mg/dL or an additional 20%) than less intensive-dose statin therapy or placebo and produced a greater reduction in CVD events. Each 1-mmol/L (38.7-mg/dL) reduction in LDL-C reduced the RR for CVD events by approximately 28%. See Table 4 for definitions of high-, moderate-, and low-intensity statin therapy. More intensive statin therapy = atorvastatin 80 mg, simvastatin 80 mg. Less intensive statin therapy = atorvastatin 10 mg, pravastatin 40 mg, or simvastatin 20-40 mg. | Н | Secondary Prevention | CTT 2010 (20)—data from 5 trials<br>TNT (46)<br>IDEAL (47)<br>PROVE-IT (48)<br>A-Z (117)<br>SEARCH (124) (not included in CQ1) |
| 12 | In trials of more intensive statin therapy (atorvastatin 80 mg, simvastatin 80 mg) compared with less intensive statin therapy (atorvastatin 10 mg, pravastatin 40 mg, or simvastatin 20–40 mg), women with CHD or acute coronary syndromes experienced a similar (approximately 25%) magnitude of relative CVD reduction as men (approximately 29%). Women also experienced a similar magnitude of absolute risk reduction as men. | Н | Secondary Prevention<br>(women included) | CTT 2010 (20)—5 trials<br>TNT (46)<br>IDEAL (47)<br>PROVE-IT (48)<br>A-Z (117)<br>SEARCH (124) (not included in CQ1) |
| 13 | In adults with and without CVD, in trials comparing more intensive to less intensive statin therapy or statin therapy with placebo/control, the relative CVD risk reduction was similar for those <65 years, 65 to ≤75, or >75 years of age. There is less information to estimate the magnitude of benefit in those under age 45 or over age 75 years, because fewer participants in these age groups were enrolled in clinical trials. More intensive statin therapy did not appear to reduce CVD risk, compared with less intensive statin therapy, in those with ASCVD and age >75 years. Statin therapy, compared with control (most RCTs evaluated moderate-intensity statin therapy), had a similar magnitude of RR reduction in those >75 as in those ≤75 years of age with and without ASCVD. Statin therapy vs. control trials = atorvastatin (A) 10-20 mg, fluvastatin (F) 80 mg, lovastatin (L) 40-80 mg, pravastatin (P) 40 mg, rosuvastatin (R) 10-20 mg, simvastatin (S) 40 mg. See Table 4 for the Expert Panel's definitions for high-, moderate-, and low-intensity statin therapy. The Panel uses <i>moderate intensity</i> to refer to statin drugs and doses that lower LDL-C by 30% to approximately 50%. This dose refers to atorvastatin 10 mg, fluvastatin 80 mg, lovastatin 40 mg, pravastatin 40 mg, pravastatin 40 mg, and simvastatin 40 mg. | H | Primary Prevention,<br>Secondary Prevention | CTT 2010 (20)—26 trials Included: More vs. less statin TNT (46) IDEAL (47) PROVE-IT (48) A-Z (117) SEARCH (124) Statin vs. control (statin/dose, percent LDL-C reduction) 4S (47) S20-40, -36% WOSCOPS (72) P40, -22% CARE (130) P40, -29% AFCAPS/TexCAPS (17) L20-40, -24% LIPID (74) P40, -27% GISSI-P (86) P20, -9% LIPS (122) F40 BID, -27% HPS (16) S40, -38% PROSPER (38) P40, -27% ALLHAT-LLT (131) P40, -14% ASCOT-LLA (132) A10, -31% ALERT (133) F40, -20% CARDS (75) A10, -38% ALLIANCE (118)—NA 4D (87)—A20, -27% ASPEN (119) A10, -34% MEGA (18) P10-20, -17% JUPITER (49) R20, -40% GISSI-HF (86) R10, -30% AURORA (84) R10, -38% |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 14 | In adults with CHD (including acute coronary syndromes, or a history of MI, stable or unstable angina, coronary revascularization), statin therapy reduced the RR for CVD events by approximately 21% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. This relationship was similar for more intensive compared with less intensive statin therapy and for statin therapy compared with placebo/control. | Н | Secondary Prevention | СТТ 2010 (20)—26 trials—see above |
| 15 | In adults with CVD other than CHD (including stroke, TIA presumed to be of atherosclerotic origin, or peripheral arterial disease or revascularization), statin therapy reduced the RR for CVD events by approximately 19% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. This relationship was similar for more intensive compared with less intensive statin therapy and for statin therapy compared with placebo/control. | н | Secondary Prevention | CΠ 2010 (20)—26 trials |
| 16 | In adults with diabetes and CHD or other CVD, moderate-dose statin therapy reduced CVD events by approximately 20% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. | н | Secondary Prevention<br>(diabetes subgroup<br>included) | CTT 2008 (134)—14 trials |
| .7 | In adults with and without CVD, statin therapy reduced CVD events in both men and women. | Н | Primary Prevention,<br>Secondary Prevention | CTT 2010 (20)—26 trials |
| 18 | In adults with and without CVD, in trials comparing more* intensive with less intensive statin therapy, or statin therapy with placebo/control, there were no clinically important differences in the CVD risk reduction between the subgroups listed below: • Treated hypertension or all others • Systolic blood pressure $<140, \ge 140$ to $<160,$ and $\ge 160$ mm Hg • Diastolic blood pressure $<80, \ge 80$ to $<90,$ and $\ge 90$ mm Hg • Body mass index $<25, \ge 25$ to $<30,$ and $\ge 30$ kg/m² • Current smoking and nonsmokers GFR $<60, 60$ to $<90, \ge 90$ mL/min per 1.73 m²) • Post-Ml • Total cholesterol $\le 5.2$ (201 mg/dL), $>5.2$ to $6.5, >6.5$ (251 mg/dL) mmol/L • Triglycerides $\le 1.4$ (124 mg/dL), $>1.4$ to $2.0, >2.0$ (177 mg/dL) mmol/L • HDL-C $\le 1.0$ (39 mg/dL), $>1.0$ to $\le 1.3, >1.3$ (50 mg/dL) mmol/L | н | Primary Prevention,<br>Secondary Prevention | CΠ 2010 (20)—26 trials |
| 9 | In more vs. less statin and statin vs. control trials combined, each 1-mmol/L $(38.7\text{-mg/dL})$ reduction in LDL-C resulted in approximately 22% reductions in CVD risk across baseline LDL-C levels [<2 mmol/L (77 mg/dL), $\geq$ 2 to <2.5 mmol/L (97 mg/dL), $\geq$ 2.5 to <3.0 mmol/L (116 mg/dL), $\geq$ 3.0 to <3.5 mmol/L (135 mg/dL), and $\geq$ 3.5 mmol/L, either untreated or on statin therapy]. In the statin vs. placebo/control trials, those with LDL-C <2 mmol/L may have experienced less benefit than those with higher LDL-C level. | М | | CΠ 2010 (20)—26 trials |
| :0 | In adults, statins reduce the RR for CVD, CHD, and fatal CHD similarly in those with or without hypertension. This benefit applies across all levels of baseline systolic and diastolic blood pressure and in those with treated hypertension. | Н | Primary Prevention,<br>Secondary Prevention | CTT 2010 (20), Messerli AJC 2008 (135) |
| 1 | In adults with and without CVD who received more intensive compared with less intensive statin therapy, or statin therapy compared with placebo/control, the RR for first stroke was reduced by approximately 16% per 1-mmol/L (38.7-mg/dL) LDL-C reduction, primarily because of an approximately 21% reduction in the RR for ischemic stroke. | M to H | Primary Prevention,<br>Secondary Prevention | CTT 2010 (20)—26 trials |
| 22 | In adults with and without CHD/CVD who received more intensive compared with less intensive statin therapy, or statin therapy compared with placebo/control: • The RR for major coronary events was reduced by approximately 24% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. • The RR for nonfatal myocardial infarction was reduced by approximately 27% per 1-mmol/L LDL-C reduction. • Total mortality was reduced by approximately 10% per 1-mmol/L (38.7-mg/dL) LDL-C reduction, primarily because of a 16% reduction in the risk for cardiac death. • The risk for CVD mortality was reduced by approximately 14% per 1-mmol/L (38-mg/dL) LDL-C reduction, primarily because of a 16% reduction in the risk for cardiac death. | н | Primary Prevention,<br>Secondary Prevention | CΠ 2010 (20)—26 trials |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 23 | In adults with CHD or acute coronary syndromes who received more intensive compared with less intensive statin therapy, the RR for coronary revascularization was reduced by approximately 34% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. | Н | Secondary Prevention | CTT 2010 (20)—5 trials |
| 4 | In adults with and without CVD who received statin therapy compared with placebo/control, the RR for coronary revascularization was reduced by approximately 24% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. | н | Primary Prevention,<br>Secondary Prevention | CTT 2010 (20)—21 trials |
| 5 | In adults with and without CVD who received statin therapy, a larger absolute reduction in LDL-C (mmol/L or mg/dL) was associated with a greater reduction in the risk for CVD. | М | Primary Prevention,<br>Secondary Prevention | CTT2010 (20), Kizer 2010 (136) |
| 6 | In adults with and without CVD who received statin therapy, there was no variation in the relative reduction of CVD risk among the trials after adjustment for LDL-C reduction. Thus, LDL-C reduction appeared to account for the reduction in CVD risk. | М | Primary Prevention,<br>Secondary Prevention | СП 2010 (20) |
| 7 | Consistent 23%-28% relative reductions in CVD risk per 39-mg/dL (1-mmol/L) reduction in LDL-C were observed after 1 year to beyond 5 years of statin treatment. | Н | Secondary Prevention,<br>Primary Prevention | CTT 2008 (134), 2005 (50) CTT 2010 (96) |
| 8 | Statins reduce the RR for CVD similarly in primary- and secondary-<br>prevention populations. | Н | Primary Prevention;<br>Secondary Prevention | CTT 2010 (20) CTT 2010 Web appendix (50) |
| 9 | In adults with diabetes (some of whom had CHD), statin therapy reduced the RR for CVD events by approximately 20% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. This 1-mmol (20%) risk-reduction relationship was similar for more intensive compared with less intensive statin therapy and for statin therapy compared with placebo/control. | н | Secondary Prevention<br>(includes diabetes<br>subgroup)<br>Primary Prevention in<br>Individuals With<br>Diabetes | CΠ 2010 (20) CΠ 2008 (134) |
| 0 | Adults with type 2, type 1, and no diabetes had similar RRRs in CVD per 1-mmol/L (38.7-mg/dL) LDL-C reduction. | Н | Primary Prevention in<br>Individuals With<br>Diabetes | СП 2010 (20) |
| 1 | In adults with diabetes without CVD, moderate-dose statin therapy, compared with placebo/control, reduced the RR for CVD events by approximately 27% per 1-mmol/L (38.7-mg/dL) LDL-C reduction. | Н | Primary Prevention in<br>Individuals With<br>Diabetes | CTT 2008 (134)—14 trials |
| 2 | In adults with diabetes, statin therapy reduced the RR for CVD by a similar magnitude for subgroups of diabetic men and women, $<65$ and $\geq65$ years of age; treated hypertension; body mass index $<25, >25$ to $<30,$ and $\geq30$ ; systolic blood pressure $<160$ and $\geq160$ mm Hg; diastolic blood pressure $<90$ and $\geq90$ mm Hg; current smokers and nonsmokers; estimated GFR $<60, \geq60$ to $<90,$ and $\geq90$ mL/min/ $1.73$ m²; and predicted annual risk for CVD $<4.5\%, >4.5\%$ to $<8.0\%,$ and $\geq8.0\%.$ Whereas RRRs are similar across these subgroups, absolute risk reductions may differ for various subgroups. | Н | Primary Prevention in<br>Individuals With<br>Diabetes | CTT 2008 (134)—14 trials |
| 3 | In adults 40 to 75 years of age with diabetes and ≥1 risk factor, fixed moderate-dose statin therapy that achieved a mean LDL-C of 72 mg/dL reduced the RR for CVD by 37% (in this trial, LDL-C was reduced by 46 mg/dL or 39%). | М | Primary Prevention in<br>Individuals With<br>Diabetes | CARDS (75) |
| 4 | In men and postmenopausal women 40 to 73 years of age without CHD/CVD, the majority of whom did not have diabetes and had baseline LDL-C levels <190 mg/dL, fixed low- to moderate-dose statin therapy that achieved a mean LDL-C of 115–127 mg/dL reduced the RR for CVD by 24%–25%, compared with placebo, with mean LDL-C levels of 153–156 mg/dL. (In these trials, LDL-C was reduced by 29–35 mg/dL and 19%–25% from baseline with a low- to moderate-dose statin.) | Н | Primary Prevention | AFCAPS (17); MEGA (18) |
| 5 | In men $\geq$ 50 years and women $\geq$ 60 years of age without CHD/CVD with LDL <130 mg/dL and hs-CRP $\geq$ 2 mg/L, fixed intensive-dose statin that achieved a mean LDL-C of 53 mg/dL reduced the RR for CVD events by 44% compared with placebo, which had a mean LDL-C 110 mg/dL. In this trial, LDL-C was reduced by 53 mg/dL, or 49%. | М | Primary Prevention | JUPITER (49) |
| 6 | In adults without CVD (some of whom had diabetes) who received more intensive or less intensive statin therapy, or statin therapy compared with placebo/control, the RR for CVD events was reduced by approximately 25% per 1-mmol/L LDL-C reduction. This was similar to the CVD RRR observed in those with CHD or CVD. | Н | Primary Prevention | СТТ 2010 (20) |
| 7 | Statin therapy reduces CHD and stroke events in adults $\geq$ 40 years of age without CHD/CVD, and with a wide range of baseline LDL-C levels. | н | Primary Prevention | CTT 2010 (20) JUPITER (49) AFCAPS (17) MEGA (18) |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 38 | Statin therapy, with a range of LDL-C lowering, reduces all-cause mortality, compared with placebo, in primary-prevention clinical trials of adults who were in general $\geq$ 40 years of age and had at least 1 risk factor, and with a wide range of baseline LDL-C levels. | M | Primary Prevention | СП 2010 (20) |
| 39 | There is insufficient evidence to determine the benefit of statins in primary prevention on all-cause mortality separately for women and men or with advancing age. | I | Primary Prevention | СП 2010 (20) |
| 40 | In MEGA (18), AFCAPS (17), JUPITER (49), and CARDS (75), the 10-year NNTs to prevent 1 hard CVD event were 82, 56, 30, and 15, respectively. These reflect RRRs of 24%, 26%, 44%, and 37%, respectively, and placebo event rates for major CVD calculated at 10 years of 5.1%, 6.9%, 7.6%, and 18%, respectively. | M | Primary Prevention | CTT 2010 (20) appendix individual trials—projected calculation |
| 41 | In adults without CVD (some of whom had diabetes) overall, who received statin therapy compared with placebo/control, the RR for CVD events was reduced by approximately 25% per 1-mmol/L LDL-C reduction. This was similar to the CVD RRR observed in those with CHD or CVD. | Н | Primary Prevention,<br>Primary Prevention in<br>Individuals With<br>Diabetes | СТТ 2010 (20) |
| 42 | Statin therapy, with a range of LDL-C lowering, reduces all-cause mortality by about 10%, compared with placebo, in primary-prevention clinical trials of adults who were ≥40 years of age and in general who had at least 1 risk factor, and with a wide range of baseline LDL-C levels. | М | Primary Prevention,<br>efficacy | Cochrane (15), Ray (137), Brugts (138),<br>Bukkapatnam (139), JUPITER (49)<br>MEGA—women (140) |
| 43 | In adults with and without CVD, intensive- and moderate-dose statins do not increase the risk for death from noncardiovascular causes, regardless of baseline LDL-C. Statins do not increase (or decrease) the risk for incident cancer overall or cancer of any type, or the risk for cancer death. | Н | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins | CTT 2010 (20), Mills 2008 (97), Cochrane (15),<br>Bonovas (141) |
| 44 | In adults with or without CVD, statin therapy is associated with an excess risk for incident diabetes. Statin therapy was associated with 1 excess case of incident diabetes per 1,000 individuals treated for 1 year, compared with placebo/control, with little heterogeneity among 13 trials (including JUPITER [49]). Risk for diabetes was highest in older persons (NNH=1,002 per year). Statin therapy resulted in 5.4 fewer major CVD events per 1-mmol/L LDL-C reduction per 1,000 individuals treated for 1 year compared with placebo (NNT to benefit, 185 per year). High-intensity statin therapy was associated with 2 excess cases of incident diabetes per 1,000 individuals treated for 1 year, compared with moderate-intensity statins (NNH=498 per year). High-intensity statin therapy resulted in 6.5 fewer major CVD events per 1,000 individuals treated for 1 year, compared with moderate-intensity statin therapy (NNT=155 per year). Rosuvastatin 20 mg was associated with 3 excess cases of incident diabetes per 1,000 individuals treated for 1 year, compared with placebo (NNH=332 per year). Rosuvastatin 20 mg resulted in 5.9 fewer major CVD events per | М | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins | Sattar 2010 (81) Preiss (142), PROVE-IT (48), A-Z (117), TNT (46), IDEAL (47), SEARCH (124), JUPITER (49) |
| | 1,000 individuals treated for 1 year, compared with placebo (NNT=169 per year). | | | |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 45 | In trials of high-intensity compared with moderate-intensity statins (clinical CVD), moderate-intensity statin compared with placebo (diabetes—primary prevention), high-intensity statin compared with placebo (secondary and primary prevention), or statin-niacin versus placebo, participants were: • Seen at visits that occurred at 4–13 weeks after randomization, and every 3–6 months thereafter. • Counseled on diet (IDEAL [47], AFCAPS [17], MEGA [18], PROVE-IT [48], SPARCL [107]) and lifestyle (JUPITER [49]) at baseline and regularly thereafter or when LDL-C increased (JUPITER [49], CARDS [75]). • Assessed for adherence to study medication at every visit. • Assessed for adverse effects by history and laboratory measurements at every visit or every other visit. | Н | Statin Adherence | Reflects review of TNT (46), IDEAL (47), PROVE-IT (48), CARDS (75), JUPITER (49), SPARCL (107), MEGA (18), AFCAPS (17) baseline and main papers; these were statin trials that demonstrated significant CVD risk reduction (and were the basis of recommendations arising from CQ1 and CQ2) HATS (121) |
| | 80 mg could be reduced to 40 mg (IDEAL [47], PROVE-IT [48]) or pravastatin 40 mg could be reduced to 20 mg (PROVE-IT [48]) or simvastatin reduced by 10 mg/d (HATS [121]). • Able to reduce the statin dose if LDL-C decreased to <39 mg/dL (1.0 mmol/L) (per investigator discretion in IDEAL [47]) or reduce the statin dose if total cholesterol was <100 mg/dL on 2 successive visits (AFCAPS [17]) or reduce by 10 mg simvastatin per day if LDL-C was <40 mg/d (HATS [121]), although they continued on study drug no matter how low the cholesterol in CARDS (75). | | | |
| | <ul> <li>Allowed to have their statin doses uptitrated or switched to more potent statin to further reduce</li> <li>LDL-C (IDEAL [47], CARDS [75], AFCAPS [17], MEGA [18], PROVE-IT [48]—pravastatin to 80 mg) if LDL-C exceeded 125 mg/dL.</li> <li>Given counseling on diet and/or glycemic control when LDL-C or triglyceride levels increased (CARDS [75]).</li> <li>Had study medication discontinued for CK ≥10 × ULN with muscle aches or weakness, or persistent ALT ≥3 × ULN on 2 consecutive tests (JUPITER [49], CARDS [75]); the dose of atorvastatin or pravastatin could be halved for abnormal LFTs, CK elevations, or myalgias (PROVE-IT [48]).</li> </ul> | | | |
| 46 | Most RCTs of moderate-intensity statin therapy and all RCTs of high-<br>intensity statin therapy excluded subjects with serious comorbidities<br>and other conditions or concomitant drug therapy predisposing to<br>adverse events from statin therapy (see Table 9). | н | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins,<br>Safety of Nonstatins | RCTs included in CQ1, 2, and 3: A-Z (117), ACCORD (14), AIM-HIGH (9), ASPEN (119), CARE (130), CDP (101), FIELD (115), GREACE (120), HATS (121), HHS (111), HPS (16), IDEAL (47), JUPITER (49), LIPID (74), LIPS (122), LRC (113), MIRACL (93), MUSHASHI-AMI (123), PROVE-IT (48), SEAS (108), SHARP (109), SPARCL (107), TNT (46) |
| 47 | In adults with and without CVD who received more intensive compared with less intensive statin therapy, or statin therapy compared with placebo/control, overall the RR for first hemorrhagic stroke was not increased. Hemorrhagic stroke comprised 11% of total strokes in the more intensive/statin group, compared with 8% in the less intensive/control groups. | М | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins | СТТ 2010 (20) |
| 48 | In adults with and without CVD, statin-treated individuals in clinical trials are not more likely to discontinue treatment than placebo-treated individuals. | Н | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins | Cochrane—14 trials (15), CTT 2010 (20) |
| 49 | In adults with and without CVD in clinical trials, low- to moderate-dose statins do not increase the risk for myalgias or muscle pain. | н | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins | Cochrane—14 trials (15), CTT 2010 (20) |
| 50 | In adults selected for participation in clinical trials of statin therapy, rhabdomyolysis occurred rarely ( $<0.06\%$ over a mean 4.8- to 5.1-year treatment period). | Н | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins | СТТ 2010 (20) |
| 51 | In adults with CHD, the rate of creatine kinase elevation $\geq$ 3 times ULN occurs infrequently and at a similar rate in those treated with intensive-or moderate-dose statin therapy. | Н | Primary Prevention,<br>Secondary Prevention,<br>Safety of Statins | Dale (98), CTT 2010 (20) |
| 52 | In adults with CHD, although uncommon (<1.5% over 5 years), intensive statin therapy increases the risk for elevated hepatic transaminase (ALT and/or AST) levels $\geq$ 2-3 times ULN more than moderate-dose statin therapy. No cases of hepatic failure were reported. | н | Primary Prevention,<br>Safety of Statins | Dale (98), Cochrane (15), CTT 2010 (20), TNT (46), IDEAL (47), PROVE-IT (48), JUPITER (49) |
| 53 | Low- to moderate-dose statin therapy has similar rates of elevated hepatic transaminase levels as placebo/no statin treatment. In general, clinical trials tend to underestimate those likely to have side effects, often related to selection procedures. | Н | Primary Prevention,<br>Safety of Statins | CTT 2010 (20) |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 54 | With the exception of simvastatin 80 mg, intensive- and moderate-dose statins did not increase the risk for rhabdomyolysis. | L | Safety of Statins | CTT 2010 (20), Cochrane (15), Mills (97) |
| 55 | In adults with CHD, CK elevation ≥3 times ULN occurs infrequently and at a similar rate in those treated with intensive- or moderate-dose statin therapy (0.02% [moderate-dose statin] to 0.1% [higher-dose statin]) over a 1- to 5-year treatment period (RR 2.63, 95% CI 0.88–7.85). | Н | Secondary Prevention,<br>Safety | Dale 2007 (98) |
| 56 | The Expert Panel did not find evidence that statins had an adverse effect on cognitive changes or risk of dementia. | I | Safety of Statins | Reviewed RCTs in CQ1, CQ2; assessment of cognitive function only reported in HPS (16) |
| 57 | In men with CHD who are 30 to 64 years of age, immediate-release niacin (with an approximately 2-g dose): • Decreased total cholesterol by 10% and triglycerides by 27%. • Markedly increased the risk for adverse skin events (including flushing, pruritus, acanthosis nigricans, and other types of skin rash). • Increased the risk for other adverse events: • Atrial fibrillation • Gastrointestinal events (including nausea, stomach pain, decreased appetite, and unexplained weight loss) • Gout • Elevated levels of uric acid, serum glutamic oxaloacetic transaminase, alkaline phosphatase, and glucose • Lipids, LFTs, uric acid, and glucose were monitored during up-titration and every 4-12 months thereafter. | L | Secondary Prevention,<br>Safety,<br>Monotherapy,<br>Safety,<br>Efficacy | CDP (101,143) |
| 58 | <ul> <li>In a trial in 67 adults with CHD and low HDL-C, slow-release niacin (at a mean 2.4-g dose) plus low-dose simvastatin resulted in the following:</li> <li>Low levels of LDL-C and raised levels of HDL-C.</li> <li>Although not powered to detect a reduction in CVD events, the rate of major clinical events was 90% lower than that in the placebo group.</li> <li>Slow-release niacin did not cause flushing in this trial.</li> <li>The simvastatin-niacin group had increased ALT, CK, uric acid, and homocysteine.</li> <li>Antioxidant vitamins diminished the beneficial effect of niacin on HDL-C.</li> <li>Lipids, LFTs, uric acid, and glucose were monitored during up-titration and every 2-4 months thereafter.</li> </ul> | L | Secondary Prevention, Combination Treatment | HATS Investigators (121) |
| 59 | In adults 45 years of age and older with established CVD and low HDL-C (<40 mg/dL in men or <50 mg/dL in women), elevated triglycerides (150-400 mg/dL), and LDL-C <180 mg/dL off statin, in whom the dose of simvastatin was adjusted, or ezetimibe was added, to maintain LDL-C in a range of 40-80 mg/dL, extended-release niacin 1,500-2,000 mg/day plus simvastatin (9.5% also on ezetimibe 10 mg) compared with placebo (with 50 mg immediate-release niacin) plus simvastatin (21.5% also on ezetimibe 10 mg: • Improved the lipid profile without a further decrease in CVD events. Specifically, it lowered LDL-C levels an additional 6%, increased HDL-C by an additional 14%, reduced triglycerides by an additional 23%, lowered apolipoprotein B by an additional 10%, and reduced lipoprotein(a) by an additional 19%. • There were similar rates of CVD events in subgroups by age, sex, or diabetes, metabolic syndrome, or previous myocardial infarction status, as well as similar rates of adverse events, including liver function abnormalities, muscle symptoms, and rhabdomyolysis. • Lipids, LFTs, uric acid, and glucose were monitored during up-titration and every 3-12 months thereafter. | M | Secondary Prevention, Combination Treatment | AIM-HIGH Investigators (9) |
| 60 | In men 35–59 years of age without CHD, hypertension, diabetes, or obesity and with LDL-C ≥175 mg/dL and triglycerides <300 mg/dL, cholestyramine: • Reduced LDL-C by 13%, with minimal changes in triglycerides or HDL-C levels. • Reduced the RR for CHD events by 19%. • Increased the risk for adverse gastrointestinal effects, including constipation, heartburn, abdominal pain, belching, bloating, gas, nausea. • Adherence was only modest. | L | Primary Prevention,<br>Safety,<br>Efficacy | LRC (113) |
| 61 | Insufficient data to evaluate the efficacy and safety of ezetimibe monotherapy. | I | Efficacy,<br>Safety,<br>Nonstatin | |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 62 | Insufficient data to evaluate the additional efficacy and safety of ezetimibe in combination with a statin compared with a statin alone. | I | Safety,<br>Efficacy,<br>Combination Treatment | |
| 3 | In adults 45–85 years of age with mild to moderate aortic stenosis and without CVD or diabetes, simvastatin 40 mg coadministered with ezetimibe 10 mg, compared with placebo: • Decreased LDL-C by an average of 50%. • Reduced the RR for CVD events by 22% over 4.35 years of treatment. • Increased the risk for elevated hepatic transaminases. | L | Safety,<br>Efficacy,<br>Combination Treatment | SEAS (108) |
| 1 | In adults ≥40 years of age with CKD, of whom 33% were receiving dialysis (peritoneal or hemodialysis), ezetimibe 10 mg coadministered with simvastatin 20 mg, compared with placebo: • Lowered LDL-C by 37 mg/dL (33%) in those who were not receiving dialysis and by 23% in those who were receiving dialysis. • Reduced the risk for CVD events by 17% overall and 21% in those without CVD. • Reduced the risk for CVD events by 22% in those who were not receiving dialysis. • Did not reduce CVD events in those with CVD or in those receiving hemodialysis. • Modestly increased the risk for muscle symptoms requiring discontinuation of treatment (1.1% vs. 0.6% with p=0.02). • Did not increase the risk for elevated hepatic transaminases, cancer, hemorrhagic stroke, or noncardiovascular mortality. | L | Safety,<br>Efficacy,<br>Combination Treatment,<br>CKD | SHARP (109) |
| 5 | Ezetimibe coadministered with simvastatin does not appear to increase the risk for cancer compared with placebo. | L | Safety,<br>Combination Treatment | SHARP (109) |
| 96 | In adults 50-75 years of age with diabetes—with total cholesterol <250 mg/dL, and total cholesterol/HDL ratio ≥4.0 or triglycerides <450 mg/dL—fenofibrate, compared with placebo: • Modestly reduced LDL-C, minimally increased HDL-C, and substantially reduced triglycerides. • In those without clinical CVD, reduced the risk for CHD/CVD events. • In those with clinical CVD, did not reduce the risk for CHD/CVD events. • Was no different than placebo for myositis or rhabdomyolysis, CK or ALT elevations, renal disease requiring hemodialysis, or cancer. • Was associated with higher rates of pancreatitis and pulmonary embolism, and increased creatinine levels on average by 0.113-0.136 mg/dL (10-12 mmol/L). | L | Safety,<br>Efficacy,<br>Nonstatin Treatment | FIELD (115) |
| 7 | In adults 40-79 years of age with diabetes, CVD, and/or CVD risk factors, with LDL-C 60-180 mg/dL, HDL-C <55 mg/dL in women and black individuals, HDL-C <50 mg/dL for all others, and triglycerides <750 mg/dL on no medication or <400 mg/dL on medication: • Fenofibrate added to simvastatin did not additionally reduce LDL-C, minimally increased HDL-C (1 mg/dL or 2%), and moderately reduced triglycerides (23 mg/dL or 14%), compared with simvastatin therapy, which had on-treatment mean LDL-C of 80 mg/dL, HDL-C of 40.5 mg/dL, and triglycerides of 170 mg/dL. • In the trial overall, and in those without and with clinical CVD, fenofibrate-simvastatin did not reduce the risk for CVD events compared with simvastatin alone. • Those with triglycerides ≥204 mg/dL and HDL-C ≤40 mg/dL may have experienced a reduction in CVD events from fenofibrate-simvastatin, compared with simvastatin alone. • Fenofibrate-simvastatin had similar rates as simvastatin alone for myopathy, myositis, or rhabdomyolysis; CK or ALT elevations, renal disease requiring hemodialysis; cancer death; or pulmonary embolism/thrombosis. • Fenofibrate-simvastatin was more likely to increase ALT >5 times ULN and to increase creatinine level. • CVD event rates were higher in women with well-controlled diabetes who received fenofibrate-simvastatin compared with simvastatin alone. | M | Safety,<br>Efficacy,<br>Nonstatin Treatment | ACCORD (14) |
| 8 | In men 40–55 years of age without CHD or CHF and non–HDL-C ≥200 mg/dL, gemfibrozil: • Reduced LDL-C by 10% and triglycerides by 43%, and increased HDL-C by 10%. • Reduced the RR for CHD by 37%, compared with placebo. • Increased skin cancer, increased gastrointestinal surgery, and increased severe upper gastrointestinal symptoms, especially in first year. There was no difference in diarrhea, constipation, nausea, or | M | Safety,<br>Efficacy,<br>Nonstatin Treatment | Helsinki Heart Study (111) |

| ES No. | Evidence Statement | Level of<br>Evidence | Recommendation(s)/<br>Section | References |
|---|---|---|---|---|
| 69 | In men with CHD who were <74 years of age with HDL-C ≤40 mg/dL and LDL-C ≤140 mg/dL, and triglycerides ≤300 mg/dL, gemfibrozil, compared with placebo: • Did not reduce LDL-C, but did reduce triglycerides by 31% and increase HDL-C by 6%. • Reduced the RR for CVD by 24%. | М | Efficacy,<br>Nonstatin Treatment | VA-HIT (114) |
| 70 | In Japanese men who were 40-75 years of age and postmenopausal women ≤75 years of age with and without CHD and LDL-C ≥170 mg/dL, EPA 1,800 mg added to statin therapy: • Did not reduce LDL-C and modestly reduced triglycerides (5%), compared with statin therapy alone. • Reduced the risk for CHD events (including revascularization and unstable angina) by 19%, compared with statin therapy alone. • Caused a similar magnitude of risk reduction in primary- and secondary-prevention populations, but the study was insufficiently powered to evaluate these populations separately. • Increased the risk for gastrointestinal disturbance, skin abnormalities, hemorrhage, and abnormal serum glutamic oxaloacetic transaminase. | М | Efficacy,<br>Safety,<br>Combination Treatment | JELIS (110) |
| 71 | In individuals with NYHA Classes II-IV systolic or ischemic heart failure, initiation of a statin did not change the absolute or RR for CVD compared with placebo. | М | Efficacy, Selected Population Subgroups | CORONA (85) from CQ1 |
| 72 | In individuals receiving maintenance hemodialysis, initiation of a statin did not change the relative or absolute risk for CVD compared with placebo. | М | Efficacy, Selected Population Subgroups | 4D (87) and AURORA (84) CQ1 & CQ2,<br>SHARP (109)—HD subgroup |
| 73 | In men and women of mean age 58 to 68 years with aortic stenosis, treatment with statin or statin plus ezetimibe for a mean of 2.1–4.4 years resulted in a reduction in LDL-C of 50%–55% (67–73 mg/dL) from a baseline LDL-C of 123–140 mg/dL and did not alter the progression of aortic stenosis as assessed by change in valve area, peak aortic valve jet velocity, peak or mean aortic valve gradient, or need for aortic valve surgery. | Н | Aortic Stenosis,<br>Combination Treatment | Parolari (144) |
| 74 | Women who were pregnant or nursing were excluded from statin, fenofibrate, niacin-statin, and ezetimibe-statin RCTs. Only men were enrolled in RCTs of niacin, BAS, and gemfibrozil. | Н | Primary Prevention,<br>Secondary Prevention | All RCTs CQ1, CQ2, and CQ3 |
| 75 | Only individuals with primary hypercholesterolemia were included in RCTs. | н | Primary Prevention,<br>Secondary Prevention | AFCAPS (17) JUPITER (49) JELIS (110) HATS (121) FIELD (115) ACCORD (14) MEGA (18) |
| 76 | In the 3 exclusively primary-prevention RCTs, low-, moderate-, and high-<br>intensity statin therapy reduced the risk for ASCVD when LDL-C levels<br>were approximately 70–130 mg/dL, 130–190 mg/dL, and 160–200<br>mg/dL. | Н | Primary Prevention | JUPITER (49)<br>MEGA (18)<br>AFCAPS (17) |
| 77 | Lipids, liver function, uric acid, and glucose tests were obtained at baseline, during up-titration, and every 2-12 months thereafter. | Н | Secondary Prevention | CDP (101) (fair) 4-12 months;<br>HATS (121) (good) 2-4 months;<br>AIM-HIGH (9) (good) 3-12 months |
| 78 | Immediate- and extended-release niacin increase cutaneous adverse effects. | M | Secondary Prevention | CDP (101), AIM-HIGH (9) (not HATS [121]—<br>SIo-Niacin) |
| 79 | When used as monotherapy or with a statin, niacin increases: Hepatic function tests. Hyperglycemia. Gastrointestinal adverse effects. Gout or increased uric acid. | H<br>M<br>M<br>M | Secondary Prevention,<br>Safety | (CDP [101], HATS [121], AIM-HIGH [9]) (CDP [101], AIM-HIGH [9]—niacin dose reduced or discontinued) (CDP [101], AIM-HIGH [9]—niacin dose reduced or discontinued) Gout (CDP [101]) Increased uric acid (HATS [121]) |
| 80 | Niacin increases the incidence of atrial fibrillation and weight loss. | L | Secondary Prevention,<br>Safety | CDP (101) (atrial fibrillation not reported in AIM-HIGH [9] or HATS [121]) |

ALT indicates alanine transaminase; ASCVD, atherosclerotic cardiovascular disease; BAS, bile acid sequestrant; BID, twice daily; CHD, coronary heart disease; CHF, congestive heart failure; CK, creatine kinase; CKD, chronic kidney disease; CVD, cardiovascular disease; EPA, eicosapentaenoic acid; GFR, glomerular filtration rate; HDL-C, high-density lipoprotein cholesterol; LDL-C, low-density lipoprotein cholesterol; LTF, liver function test; MI, myocardial infarction; NNH, number needed to harm; NNT, number needed to treat; NYHA, New York Heart Association; RCT, randomized controlled trial; RR, relative risk reduction; TIA, transient ischemic attack; and ULN, upper limit of normal.

#### Appendix 5. Expanded Discussion of What's New in the Guideline

#### Focus on ASCVD Risk Reduction: 4 Statin Benefit Groups

2932

- The 2013 guideline focuses on treatment of blood cholesterol to reduce ASCVD risk. Each Expert Panel was limited in the number of CQs it could choose. When the CQs from the Risk Assessment and Lifestyle Work Groups were combined with the 3 Cholesterol Panel CQs, there were 8 CQs in total that were systematically reviewed. All 3 CQs of the Cholesterol Panel evaluated evidence from RCTs with ASCVD outcomes. CQ1 and CQ2 evaluated the evidence for LDL-C and non-HDL-C goals in secondary and primary prevention. CQ3 was a comprehensive evaluation of the reduction in ASCVD events and safety for each of the cholesterol-lowering drugs available in the United States.
- The systematic review of evidence from the highest-quality RCTs with ASCVD outcomes identified strong evidence to indicate who should get which therapy at what intensity.
- The statin RCTs provided the most extensive evidence for the greatest magnitude of ASCVD event reduction, with the best margin of safety.
- Four statin benefit groups were identified, in which the potential for an ASCVD risk-reduction benefit clearly exceeds the potential for adverse effects in:
  - 1. Individuals with clinical ASCVD
  - 2. Individuals with primary elevations of LDL-C ≥190 mg/dL
  - 3. Individuals 40-75 years of age with diabetes but without clinical ASCVD and LDL-C 70-189 mg/dL
  - 4. Individuals 40-75 years of age without diabetes or clinical ASCVD with LDL-C 70-189 mg/dL and an estimated 10-year ASCVD risk of 7.5% or higher. This requires a clinician-patient discussion.
- Because few trials have been performed with nonstatin cholesterol-lowering drugs in the statin era, and those that have been performed were unable to
  demonstrate significant additional ASCVD event reductions in the RCT populations studied, there was less evidence to support the use of nonstatin drugs for
  ASCVD prevention.
- It is difficult to determine how observational data could override the conclusions from the extensive body of evidence from the statin RCTs and the paucity of evidence from nonstatin RCTs. Inherent biases of observational data are well understood and include biases in the decisions on whom to treat and who is adherent to therapy, as well as multiple measurement biases, including verification of statin use, type and dose of statin used, consistency of use over time, and outcome ascertainment. All of these problems are addressed in intent-to-treat analyses of RCTs, which is why the FDA requires well-designed RCTs to determine drug efficacy for ASCVD event reduction and common adverse effects.
- . Other approaches to treatment of blood cholesterol have been advocated, including:
  - A. Treat to target—This strategy has been the most widely used in the past 15 years, but there are 3 problems with this approach. First, current clinical trial data do not indicate what the target should be. Second, we do not know the magnitude of additional ASCVD risk reduction that would be achieved with one target lower than another. Third, this strategy does not take into account potential adverse effects from statin monotherapy or from multidrug therapy that might be needed to achieve a specific goal. Thus, in the absence of these data, this approach is less useful than it appears (Section 3). It is possible that future clinical trials may provide information warranting reconsideration of this strategy.
  - B. Lowest is best—This approach was not taken because it does not consider the potential adverse effects of multidrug therapy with an unknown magnitude of ASCVD event reduction. Ongoing RCTs of new LDL-C-lowering drugs in the setting of maximal statin therapy may address this question.
- C. Treat level of ASCVD risk—A modified version of this approach was taken, which considers both the ASCVD risk-reduction benefits and the adverse effects of statin treatment on the basis of an extensive body of RCT evidence to determine the 4 statin benefit groups. By focusing treatment on the 4 statin benefit groups, the approach is practical and simpler to implement than the past strategies. There are also important exceptions for routine initiation of statin treatment for individuals requiring hemodialysis or with NYHA class II to IV heart failure.
- D. Lifetime risk—Treatment strategies based on lifetime ASCVD risk are problematic because of the lack of data on the long-term follow-up of RCTs >15 years, the safety and ASCVD event reduction when statins are used for periods >10 years, and treatment of individuals <40 years of age.

#### A New Perspective on LDL-C and/or Non-HDL-C Goals

- The difficulty of giving up the treat-to-goal paradigm was deliberated extensively over a 3-year period. Many clinicians use targets such as LDL-C <70 mg/dL and LDL-C <100 mg/dL for secondary and primary ASCVD prevention (non-HDL-C targets are 30 mg/dL higher). However, the RCT evidence clearly shows that ASCVD events are reduced by using the maximum-tolerated statin intensity in those groups shown to benefit. After a comprehensive review, no RCTs were identified that titrated drug therapy to specific LDL-C or non-HDL-C goals to improve ASCVD outcomes. However, one RCT was identified that showed no additional ASCVD event reduction from the addition of nonstatin therapy to further treat non-HDL-C levels once an LDL-C goal was reached. In AIM-HIGH (9), the additional reduction in non-HDL-C levels [as well as additional reductions in Apo B, Lp(a), and triglycerides in addition to HDL-C increases] with niacin therapy DID NOT further reduce ASCVD risk in individuals treated to LDL-C levels of 40-80 mg/dL.
- Use of LDL-C targets may result in under treatment with evidence-based statin therapy or overtreatment with nonstatin drugs that have not been shown to reduce
  ASCVD events in RCTs (even though the drug may additionally lower LDL-C and/or non-HDL-C). Implications of treating to an LDL-C goal may mean that a
  suboptimal intensity of statin is used because the goal has been achieved, or that adding a nonstatin therapy to achieve a specific target results in down-titration of
  the evidence-based intensity of statin for safety reasons. However, when RCT evidence is available that a nonstatin therapy further reduces ASCVD events when
  added to statin therapy, the nonstatin therapy may be considered.
- Some examples comparing a strategy based on the 4 statin benefit groups to a strategy using LDL-C/non-HDL-C targets:
- A. Secondary prevention—Evidence supports high-intensity statin therapy for this group to maximally lower LDL-C. It does not support the use of an LDL-C target. For example, if a secondary-prevention patient achieves an LDL-C of 78 mg/dL on a dose of 80 mg of atorvastatin, he/she is receiving evidence-based therapy. As of yet, there are no data to show that adding nonstatin drug(s) to high-intensity statin therapy will provide incremental ASCVD risk-reduction benefit with an acceptable margin of safety. Indeed, AIM-HIGH (9) demonstrated the futility of adding niacin in individuals with low HDL-C and high triglycerides, and ACCORD (14) demonstrated the futility of adding fenofibrate in persons with diabetes. Although an ACCORD subgroup analysis of those with high triglycerides and low HDL-C levels suggested that fenofibrate may reduce ASCVD events in patients with diabetes, this is hypothesis generating and needs further testing in comparison to the evidence-based use of a high-intensity statin. In addition, not having a goal of <70 mg/dL for LDL-C means that the patient who is adhering to optimal lifestyle management and receiving a high-intensity statin avoids additional, non-evidence-based therapy just because his/her LDL-C is higher than an arbitrary cutpoint. Indeed, the LDL-C goal approach can make this patient unnecessarily feel like a failure.

- B. Familial hypercholesterolemia with LDL-C ≥190 mg/dL—In many cases, individuals with familial hypercholesterolemia are unable to achieve an LDL-C goal <100 mg/dL. For example, an individual with familial hypercholesterolemia may achieve an LDL-C of only 120 mg/dL despite use of 3 cholesterol-lowering drugs. Although this patient may have fallen short of the 100-mg/dL goal, he/she has decreased his/her LDL-C by >50% (starting from an untreated LDL-C level of ~325-400 mg/dL). These patients are not treatment failures, as observational data has shown significant reductions in ASCVD events without achieving specific LDL-C targets. This is an area where observational data supports the recommended approach.
- C. Type 2 diabetes—For those 40-75 years of age with risk factors, the potential benefits of LDL-C lowering with a high-intensity statin are substantial. Because those with diabetes often have lower LDL-C levels than those without diabetes, "goal"-directed therapy often encourages use of a lower statin dose than is supported by the RCTs, and nonstatin drugs may be added to address low HDL-C or high triglycerides, for which RCT evidence of an ASCVD event reduction is lacking. Giving a maximally tolerated statin intensity should receive primary emphasis because it most accurately reflects the data that statins reduce the relative risk of ASCVD events similarly in individuals with and without diabetes, and in primary and secondary prevention in those with diabetes, along with evidence that high-intensity statins reduce ASCVD events more than moderate-intensity statins.
- D. Estimated 10-year ASCVD risk ≥7.5%—Data have shown that statins used for primary prevention have substantial ASCVD risk-reduction benefits across the range of LDL-C levels of 70–189 mg/dL. Moreover, the Cochrane meta-analysis (15), as well as a meta-analysis by the Cholesterol Treatment Trialists (13), confirms that primary prevention with statins reduces total mortality as well as nonfatal ASCVD events.
- RCTs are used to identify those who are unlikely to benefit from initiation of statin therapy despite being at high ASCVD risk, such as those with higher NYHA classes
  of heart failure or those on hemodialysis.

#### **Global Risk Assessment for Primary Prevention**

- . Use of the new Pooled Cohort Equations is recommended to estimate 10-year ASCVD risk in both white and black men and women who do not have clinical ASCVD.
- . By more accurately identifying higher-risk individuals for statin therapy, the guideline focuses statin therapy on those most likely to benefit.
- It also indicates, on the basis of RCT data, those high-risk groups that might not benefit. The Expert Panel emphasizes that the guideline is "patient centered" in primary prevention. It is recommended that the potential for an ASCVD risk-reduction benefits, adverse effects, and drug-drug interactions, along with patient preferences, must be considered before statins are initiated for the primary prevention of ASCVD. Other factors such as LDL-C ≥160 mg/dL may also be considered. This gives clinicians and patients the opportunity for input into treatment decisions rather than a simplistic "one-treatment-fits-all" approach to drug therapy.
- These guidelines are not a replacement for clinical judgment; they are meant to guide and inform decision making.
- Some worry that a person 70 years of age without other risk factors will receive statin treatment on the basis of age alone. The estimated 10-year risk is still ≥7.5%,
  a risk threshold for which a reduction in ASCVD risk events has been demonstrated in RCTs. Most ASCVD events occur after age 70 years, giving individuals ≥70
  years of age the greatest potential for absolute risk reduction.
- Some have proposed using selected inclusion criteria from RCTs to determine the threshold for statin initiation. However, the Cholesterol Treatment Trialists individual-level meta-analysis showed that statin therapy reduces ASCVD events regardless of categorical risk factors in both primary and secondary prevention. Therefore, the rationale for using fixed cutpoints to determine whether statin therapy should be initiated is refuted by a consideration of the total body of evidence from RCTs.
- In addition, a trial-based strategy identifies those at increased ASCVD risk less accurately than does a strategy based on an assessment of global ASCVD risk. This
  selective use of inclusion criteria excludes well-established risk factors, such as smoking and advancing age (the strongest risk factor because it represents
  cumulative risk factor exposure).
- The poor discrimination of RCT inclusion criteria for identifying those at increased 10-year ASCVD risk is shown by a calculation performed by the Risk Assessment Work Group using nationally representative data from NHANES. Use of the RCT inclusion criteria (from RCTs that found a reduction in ASCVD events to guide initiation of statin therapy) would result in the treatment of 16% of individuals with <2.5% estimated 10-year ASCVD risk and 45% of those with 2.5% to <5% estimated 10-year ASCVD risk (many would say inappropriately), whereas 38% of those with ≥7.5% 10-year ASCVD risk would not have been identified as candidates for statin therapy.

#### Safety

- RCTs are used to identify important safety considerations in individuals receiving treatment of blood cholesterol to reduce ASCVD risk and to determine statin
  adverse effects to facilitate understanding of the net benefit from statin therapy.
- Safety issues that are uncommon or unlikely to be seen in the populations studied in RCTs require more than analyses of single RCTs. This limitation was overcome,
  in part, by considering high-quality systematic reviews and meta-analyses of statin RCTs.
- Expert guidance is provided on management of statin-associated adverse effects, including muscle symptoms.
- This guideline emphasizes the importance of using additional sources of information on safety, including FDA reports, manufacturers' prescribing information, and
  pharmacists, to aid in the safe use of cholesterol-lowering drug therapy.

#### Role of Biomarkers and Noninvasive Tests

- There is a concern about other factors that may indicate elevated ASCVD risk but were not included in the Pooled Cohort Equations for predicting 10-year ASCVD risk.
- The Risk Assessment Work Group has performed an updated systematic review of nontraditional risk factors, such as CAC, and has included recommendations to
  consider their use to the extent that the evidence allows.
- In selected individuals who are not in 1 of the 4 statin benefit groups, and for whom a decision to initiate statin therapy is otherwise unclear, additional factors may be considered to inform treatment decision making.
- These factors include primary LDL-C ≥160 mg/dL or other evidence of genetic hyperlipidemias; family history of premature ASCVD with onset <55 years of age in a first-degree male relative or <65 years of age in a first-degree female relative; high-sensitivity C-reactive protein ≥2 mg/L; CAC score ≥300 Agatston units or ≥75th percentile for age, sex, and ethnicity; ankle-brachial index <0.9; and elevated lifetime risk of ASCVD. Additional factors may be identified in the future.</li>

2934

#### Future Updates to the Blood Cholesterol Guideline

- This guideline focuses on treatments proven to reduce ASCVD events. It is not and was never intended to be a comprehensive approach to lipid management.
- Using RCT evidence assessed for quality provides a strong foundation for treatment of blood cholesterol to reduce ASCVD risk that can be used now. There are many
  clinical questions for which there is an absence of RCT data available to develop high-quality, evidence-based recommendations. For these questions, expert opinion
  may be helpful to clinicians and could be developed in the next iteration of the guideline.
- . CQs for future guidelines could examine:
  - 1. the treatment of hypertriglyceridemia;
  - 2. the use of non-HDL-C in treatment decision making;
  - 3. whether on-treatment markers such as Apo B, Lp(a), or LDL particles are useful for guiding treatment decisions;
  - 4. the best approaches to using noninvasive imaging for refining risk estimates to guide treatment decisions;
  - 5. how lifetime ASCVD risk should be used to inform treatment decisions and the optimal age for initiating statin therapy to reduce lifetime risk of ASCVD;
  - 6. subgroups of individuals with heart failure or undergoing hemodialysis who might benefit from statin therapy;
  - 7. long-term effects of statin-associated new-onset diabetes and management;
  - 8. efficacy and safety of statins in patient groups excluded from RCTs to date (e.g., those who are HIV positive or have received a solid organ transplant); and
  - 9. role of pharmacogenetic testing.

AIM-HIGH indicates Atherothrombosis Intervention in Metabolic Syndrome With Low HDL/High Triglycerides and Impact on Global Health Outcomes; ACCORD, Action to Control Cardiovascular Risk in Diabetes; Apo B, apolipoprotein B; ASCVD, atherosclerotic cardiovascular disease; CAC, coronary artery calcium; CQ, critical question; FDA, U.S. Food and Drug Administration; HDL-C, high-density lipoprotein cholesterol; LDL-C, low-density lipoprotein cholesterol; LDL-C, l

<sup>\*</sup>For additional information, see http://www.mesa-nhlbi.org/CACReference.aspx.

Protocol 747-209 Version 4: 19 Dec 2016

# APPENDIX B. GUIDANCE FOR ELEVATED LIVER BIOCHEMISTRY VALUES

For subjects who progress to cirrhosis and decompensation while participating in the study, elevation in liver biochemistry and development of other laboratory and clinical abnormalities may be expected. Clinical adverse events (AEs) should be reported and recorded as described in Section 12.1.5 and appropriate action should be taken regarding investigational product use and study participation as described in Section 8.4.

However, if these abnormalities are not consistent with the pattern of change attributable to disease progression (as assessed by the Investigator) and no other cause is readily apparent (eg, acute biliary obstruction caused by gallstones in the common bile duct), further actions are appropriate as outlined below. The Sponsor should be contacted to discuss the case further.

Per guidance from the FDA (FDA 2009), subjects with normal ALT/AST and bilirubin at baseline, an increase in ALT/AST to >3× ULN or total bilirubin >2× ULN should be followed by repeat testing within 48 to 72 hours of the serum chemistry to confirm the abnormalities and to determine if they are increasing or decreasing. In conjunction with this, a physical exam should be performed and AE information should be collected. If symptoms persist or repeat testing shows ALT/AST >3× ULN or total bilirubin >2× ULN, subjects should be closely monitored. In subjects with abnormal ALT/AST or bilirubin at baseline, fold increase should be assessed against baseline levels instead of ULN as follows: 3× baseline ALT/AST, or total bilirubin >2× baseline (and >2 mg/dL). In subjects with abnormal values at baseline who develop a nadir value during the study, the reference points noted above should be changed from baseline to the nadir value for subsequent assessments.

In subjects who are far from their study site, it may be difficult for the subjects to return to the site promptly. In this case, the subjects should be retested locally, but normal laboratory ranges should be recorded, results should be made available to the Investigator immediately, and the data should be included in the case reports. If symptoms persist or repeat testing shows persistent abnormality as described above, it is appropriate to initiate close observation (defined below) to determine whether the abnormalities are improving or worsening.

If close observation is not possible, investigational product should be interrupted until further investigation can be performed.

Close observation may include:

- Repeating liver enzyme and serum bilirubin tests 2 or 3 times weekly. Frequency of retesting can decrease to once a week or less if abnormalities stabilize or the investigational product has been discontinued and the subject is asymptomatic.
- Obtaining a more detailed history of symptoms and prior or concurrent diseases.
- Obtaining a history of concomitant drug use (including nonprescription medications and herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets.
- Ruling out acute viral hepatitis types A, B, C, D, and E; autoimmune or alcoholic hepatitis; hypoxic/ischemic hepatopathy; and other biliary tract disease.

Protocol 747-209 Version 4: 19 Dec 2016

- Obtaining a history of exposure to environmental chemical agents.
- Obtaining additional tests to evaluate liver function, as appropriate (eg, INR, direct bilirubin).

Discontinuation of treatment should be considered if the following abnormality or group of abnormalities occur (in subjects with baseline values within the normal range):

- ALT or AST >8× ULN
- ALT or AST  $>5 \times$  ULN for more than 2 weeks
- ALT or AST  $>3 \times$  ULN and total bilirubin  $>2 \times$  ULN or INR >1.5)
- ALT or AST >3× ULN with the appearance of new onset fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)

In subjects with abnormal baseline values, the reference point should be changed from ULN to baseline. In subjects with abnormal values at baseline who develop a nadir value during the study, the reference points noted above should be changed from ULN or baseline to the nadir value for subsequent assessments. Baseline is defined as the average of all on-study, predose values (including Screening Visit and Day 1). A nadir value is defined as the average of at least 2 consecutive post-baseline assessments, including the lowest value, regardless of when it occurs (ie, on or off treatment). Repeat and unscheduled visits will be included in the determination of the nadir value. A new nadir value may develop over the course of the study if liver biochemistries improve over time.

Protocol 747-209 Version 4: 19 Dec 2016

# APPENDIX C. COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS

# Common Terminology Criteria for Adverse Events (CTCAE)

Version 4.0

Published: May 28, 2009 (v4.03: June 14, 2010)

#### U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES

National Institutes of Health National Cancer Institute

# Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

Publish Date: May 28, 2009

#### **Quick Reference**

The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

#### **Components and Organization**

#### SOC

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### **CTCAE Terms**

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may <u>not</u> be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

#### **Definitions**

A brief definition is provided to clarify the meaning of each AE term.

#### Grades

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

- Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL\*.
- Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.
- Grade 4 Life-threatening consequences; urgent intervention indicated.
- Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

#### Grade 5

Grade 5 (Death) is not appropriate for some AEs and therefore is not an option.

#### Activities of Daily Living (ADL)

\*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

\*\*Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

<sup>†</sup> CTCAE v4.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.com).

## CONTENTS

| SOC | Page |
|---------------------------------------------------------------------|------|
| Blood and lymphatic system disorders | 3 |
| Cardiac disorders | 4 |
| Congenital, familial and genetic disorders | 7 |
| Ear and labyrinth disorders | 8 |
| Endocrine disorders | 9 |
| Eye disorders | 10 |
| Gastrointestinal disorders | 12 |
| General disorders and administration site conditions | 22 |
| Hepatobiliary disorders | 24 |
| Immune system disorders | 26 |
| Infections and infestations | 27 |
| Injury, poisoning and procedural complications | 34 |
| Investigations | 41 |
| Metabolism and nutrition disorders | 44 |
| Musculoskeletal and connective tissue disorders | 46 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 50 |
| Nervous system disorders | 51 |
| Pregnancy, puerperium and perinatal conditions | 56 |
| Psychiatric disorders | 57 |
| Renal and urinary disorders | 59 |
| Reproductive system and breast disorders | 61 |
| Respiratory, thoracic and mediastinal disorders | 65 |
| Skin and subcutaneous tissue disorders | 71 |
| Social circumstances | 75 |
| Surgical and medical procedures | 76 |
| Vascular disorders | 77 |

| | В | lood and lymphatic syste | em disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Anemia | Hemoglobin (Hgb) <lln -="" 10.0<br="">g/dL; <lln -="" -<br="" 6.2="" <lln="" l;="" mmol="">100 g/L</lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | red by an reduction in the amount on, palpitations of the heart, soft syst | • | • • • | ay include pallor of the skin and m | ucous |
| Bone marrow hypocellular | Mildly hypocellular or <=25% reduction from normal cellularity for age | Moderately hypocellular or >25 -<br><50% reduction from normal<br>cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer than 2 weeks | Death |
| Definition: A disorder characteriz | ed by the inability of the bone mar | row to produce hematopoietic eler | ments. | | |
| Disseminated intravascular coagulation | - | Laboratory findings with no bleeding | Laboratory findings and bleeding | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by systemic pathological activated by systemic pathological activated set by systemical and coagulated by systemical pathological activation and some set of the systemical pathological activation and systemical pathological activation and systemical pathological activation and systemical pathological activation and systemical pathological activation and systemical pathological activation activation and systemical activation activatio | <del>-</del> | which results in clot formation thro | oughout the body. There is an incr | ease in the |
| Febrile neutropenia | - | - | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour. | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz degrees F) for more than one ho | ed by an ANC <1000/mm3 and a sour. | single temperature of >38.3 degre | es C (101 degrees F) or a sustain | ed temperature of >=38 degrees C | C (100.4 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and >=2 gm decrease in hemoglobin. | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate widespread erythrocyte ce | Il membrane destruction. | 1 | 1 |
| Hemolytic uremic syndrome | Evidence of RBC destruction (schistocytosis) without clinical consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder characteriz | ed by a form of thrombotic microa | ngiopathy with renal failure, hemol | lytic anemia, and severe thromboo | ytopenia. | |
| Leukocytosis | - | - | >100,000/mm3 | Clinical manifestations of leucostasis; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate an increased number of wh | nite blood cells in the blood. | | |
| Lymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz Spleen disorder | Incidental findings (e.g., Howell-Jolly bodies); mild degree of thrombocytosis and leukocytosis | Prophylactic antibiotics indicated | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder of the splee | | '<br>I | '<br> | '<br> | <u>'</u> |
| Thrombotic thrombocytopenic purpura | Evidence of RBC destruction (schistocytosis) without clinical consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | ted by the presence of microangion ual disturbances. It is an acute or s | <u>-</u> | cytopenic purpura, fever, renal abr | normalities and neurological abnor | malities such |
| Blood and lymphatic system disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | Τ | Grade | T | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute coronary syndrome | - | Symptomatic, progressive angina; cardiac enzymes normal; hemodynamically stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>unstable | Death |
| | ed by signs and symptoms related unstable angina to myocardial infa | • | lium secondary to coronary artery | disease. The clinical presentation | covers a |
| Aortic valve disease | Asymptomatic valvular | Asymptomatic; moderate | Symptomatic; severe | Life-threatening consequences; | Death |
| | thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | regurgitation or stenosis by imaging | regurgitation or stenosis by imaging; symptoms controlled with medical intervention | urgent intervention indicated (e.g., valve replacement, valvuloplasty) | |
| Definition: A disorder characteriz | ed by a defect in aortic valve funct | tion or structure. | | | |
| Asystole | Periods of asystole; non-urgent medical management indicated | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia without cardia | ac electrical activity. Typically, this | is accompanied by cessation of the | he pumping function of the heart. | |
| Atrial fibrillation | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz originates above the ventricles. | ed by a dysrhythmia without disce | rnible P waves and an irregular ve | entricular response due to multiple | reentry circuits. The rhythm distur | bance |
| Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz atria. | ed by a dysrhythmia with organize | ed rhythmic atrial contractions with | a rate of 200-300 beats per minut | te. The rhythm disturbance origina | tes in the |
| Atrioventricular block complete | - | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with complete | e failure of atrial electrical impulse | conduction through the AV node t | to the ventricles. | |
| Atrioventricular block first degree | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | - | - | - |
| | ed by a dysrhythmia with a delay i interval greater than 200 milliseco | • | tion of an electrical impulse throug | gh the atrioventricular (AV) node b | eyond 0.2 |
| Cardiac arrest | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by cessation of the pumping fu | nction of the heart. | T | 1 | 1 |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting instrumental ADL | Pain at rest; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by substernal discomfort due to | insufficient myocardial oxygenati | on. | T | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by pathological irregularities in | the cardiac conduction system. | Τ | T | |
| Constrictive pericarditis | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| Definition: A disorder characteriz | ed by a thickened and fibrotic peri | cardial sac; these fibrotic changes | impede normal myocardial function | on by restricting myocardial muscl | e action. |
| Heart failure | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences; urgent intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) | Death |
| Definition: A disorder characterize in the filling pressure. | ed by the inability of the heart to p | ump blood at an adequate volume | e to meet tissue metabolic requirer | ments, or, the ability to do so only | at an elevatior |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | Г | Grade | Г | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Left ventricular systolic dysfunction | - | - | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | ed by failure of the left ventricle to<br>nea, orthopnea, and other signs ar | | an increase in distending pressure stion and edema. | e and in end-diastolic volume. Clin | ical |
| Mitral valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in mitral valve funct | ion or structure. | | | |
| Mobitz (type) II atrioventricular block | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with relatively<br>atrioventricular (AV) node to the ve | · | block of an atrial impulse. This is the | ne result of intermittent failure of a | trial electrical |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with a progre<br>on through the atrioventricular (AV | | or to the blocking of an atrial impu | lse. This is the result of intermitter | nt failure of |
| Myocardial infarction | - | Asymptomatic and cardiac<br>enzymes minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences; hemodynamically unstable | Death |
| Definition: A disorder characteriz | ed by gross necrosis of the myoca | rdium; this is due to an interruptio | n of blood supply to the area. | | |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences; urgent intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) | Death |
| Definition: A disorder characteriz | ed by inflammation of the muscle | tissue of the heart. | T | ı | ı |
| Palpitations | Mild symptoms; intervention not indicated | Intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by an unpleasant sensation of | rregular and/or forceful beating of | the heart. | | I |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical management indicated | IV medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically; cardioversion<br>indicated | Death |
| Definition: A disorder characteriz originates in the atria. | ed by a dysrhythmia with abrupt o | nset and sudden termination of at | rial contractions with a rate of 150- | 250 beats per minute. The rhythm | disturbance |
| Pericardial effusion | - | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by fluid collection within the per | ricardial sac, usually due to inflam | mation. | <b>.</b> | I |
| Pericardial tamponade | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an increase in intrapericardi | al pressure due to the collection o | f blood or fluid in the pericardium. | Т | |
| Pericarditis | Asymptomatic, ECG or physical findings (e.g., rub) consistent with pericarditis | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic consequences (e.g., pericardial constriction) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by irritation to the layers of the | pericardium (the protective sac ar | ound the heart). | | |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences; urgent intervention indicated (e.g., valve replacement, valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in pulmonary valve | function or structure. | Ι | T | |
| Restrictive cardiomyopathy | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | ed by an inability of the ventricles | - | 1 | | |
| Right ventricular dysfunction | Asymptomatic with laboratory (e.g., BNP [B-Natriuretic Peptide ]) or cardiac imaging abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening consequences; urgent intervention indicated (e.g., ventricular assist device); heart transplant indicated | Death |
| | ed by impairment of right ventricul | | | 1 | |
| Sick sinus syndrome | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with alternation | ng periods of bradycardia and atria | 1 | ncope, fatigue and dizziness. | |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, medical intervention indicated | Severe, medically significant, medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate less than 60 beats per minute | that originates in the sinus node. | T | |
| Sinus tachycardia | Asymptomatic, intervention not indicated | Symptomatic; non-urgent medical intervention indicated | Urgent medical intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per min | nute that originates in the sinus no | de. | T |
| Supraventricular tachycardia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per min | nute that originates above the vent | tricles. | T |
| Tricuspid valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis; symptoms controlled with medical intervention | Life-threatening consequences; urgent intervention indicated (e.g., valve replacement, valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in tricuspid valve fu | nction or structure. | T | T | T |
| Ventricular arrhythmia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia that originate | s in the ventricles. | Τ | T | I |
| Ventricular fibrillation | - | - | - | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz ventricles. | ed by a dysrhythmia without disce | rnible QRS complexes due to rapi | d repetitive excitation of myocardia | al fibers without coordinated contra | action of the |
| Ventricular tachycardia | - | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates distal to the bu | ındle of His. | |
| Wolff-Parkinson-White syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically or controlled with procedure | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of an accesso | ry conductive pathway between th | e atria and the ventricles that caus | ses premature ventricular activatio | n. |
| Cardiac disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Congenital, familial and genetic disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Congenital, familial and genetic disorders - Other, specify | j , | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Ear and labyrinth dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteria | zed by a sensation of marked disco | mfort in the ear. | _ | | |
| External ear inflammation | External otitis with erythema or dry desquamation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis; stenosis or osteomyelitis; necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder characteria | zed by inflammation, swelling and r | edness to the outer ear and ear ca | anal. | • | |
| External ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | mfort in the external ear region. | _ | <b>,</b> | |
| Hearing impaired Definition: A disorder characteri | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: subjective change in hearing in the absence of documented hearing loss. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 8 kHz in at least one ear. | contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 4 kHz and above in at least one ear. | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated. Adults not enrolled in Monitoring Program: hearing loss with hearing aid or intervention indicated; limiting self care ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing aids; threshold shift >20 dB at 3 kHz and above in at least one ear; additional speech-language related services indicated. | Pediatric: Audiologic indication for cochlear implant and additional speech-language related services indicated. | |
| Middle ear inflammation | Serous otitis | Serous otitis, medical intervention indicated | Mastoiditis; necrosis of canal soft tissue or bone | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ।<br>zed by inflammation (physiologic re | ı | 1 | | 1 |
| Tinnitus | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteria | zed by noise in the ears, such as ri | nging, buzzing, roaring or clicking. | Τ | Г | |
| Vertigo | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri vertigo). | zed by a sensation as if the externa | al world were revolving around the | patient (objective vertigo) or as if | he himself were revolving in space | e (subjective |
| Vestibular disorder | - | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by dizziness, imbalance, nause | ea, and vision problems. | T | Г | |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Endocrine disord | lers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adrenal insufficiency Definition: A disorder that occurs | Asymptomatic; clinical or diagnostic observations only; intervention not indicated swhen the adrenal cortex does not | Moderate symptoms; medical intervention indicated | Severe symptoms; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | on's disease or primary adrenal ins | · - | cortisor and in some cases, the no | imone aldosterone. It may be due | to a disorder |
| Cushingoid | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms, medical intervention or hospitalization indicated | - | - |
| Definition: A disorder characterizosteoporosis, usually due to exo | zed by signs and symptoms that re genous corticosteroids. | semble Cushing's disease or synd | Irome: buffalo hump obesity, striat | ions, adiposity, hypertension, diab | etes, and |
| Delayed puberty | - | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age<br>14 yrs for females; no increase<br>in testes volume or no Tanner<br>Stage 2 by age 16 yrs for<br>males; hormone replacement<br>indicated | - | - |
| Definition: A disorder characterize | zed by unusually late sexual maturi | ty. | | | |
| Growth accelerated | - | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | - | - | - |
| Definition: A disorder characterize | zed by greater growth than expecte | ed for age. | T | T | 1 |
| Hyperparathyroidism | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characterize the blood). | zed by an increase in production of | parathyroid hormone by the para | thyroid glands. This results in hype | ercalcemia (abnormally high levels | of calcium in |
| Hyperthyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid suppression therapy indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by excessive levels of thyroid h | ormone in the body. Common car | uses include an overactive thyroid | gland or thyroid hormone overdos | e. |
| Hypoparathyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; medical intervention or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by a decrease in production of | parathyroid hormone by the parat | hyroid glands. | | |
| Hypothyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid replacement indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a decrease in production of | | and.<br>T | | |
| Precocious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical markers of puberty for females <8 years and males <9 years | - | - | - |
| Definition: A disorder characteriz 9 for boys. | zed by unusually early developmen | t of secondary sexual features; th | e onset of sexual maturation begir | ns usually before age 8 for girls an | d before age |
| Virilization | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | zed by inappropriate masculinization | n occurring in a female or prepub | ertal male. | | |
| Endocrine disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Eye di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Blurred vision | Intervention not indicated | Symptomatic; limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by visual perception of u | nclear or fuzzy images. | 1 | I | 1 |
| Cataract | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | (20/40 or better) | Symptomatic with marked decrease in visual acuity (worse than 20/40 but better than 20/200); operative intervention indicated (e.g., cataract surgery) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder chara:<br>untreated. | cterized by partial or complete op | eacity of the crystalline lens of o | one or both eyes. This results in | n a decrease in visual acuity an | id eventual blindness if |
| Conjunctivitis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; topical intervention indicated (e.g., antibiotics); limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by inflammation, swelling | g and redness to the conjunctiv | ra of the eye. | Γ | |
| Corneal ulcer | - | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Limiting self care ADL;<br>declining vision (worse than<br>20/40 but better than 20/200) | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | - |
| Definition: A disorder charac | cterized by an area of epithelial to | ssue loss on the surface of the | cornea. It is associated with in | flammatory cells in the cornea | and anterior chamber. |
| Dry eye | Asymptomatic; clinical or diagnostic observations only; mild symptoms relieved by lubricants | instrumental ADL | Decrease in visual acuity (<20/40); limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by dryness of the cornea | 1 | | | <u> </u> |
| Extraocular muscle paresis | Asymptomatic; clinical or diagnostic observations only | 1 | Limiting self care ADL; disabling | - | - |
| | cterized by incomplete paralysis | | | | |
| Eye pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | cterized by a sensation of marked | 1 | | | <u> </u> |
| Eyelid function disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | limiting instrumental ADL | Limiting self care ADL;<br>operative intervention<br>indicated | - | - |
| | cterized by impaired eyelid functi | | | | <u> </u> |
| Flashing lights | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by a sudden or brief burs | 1 | T | | T |
| Floaters | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by an individual seeing s | i | | | or or lens. |
| Glaucoma | Elevated intraocular<br>pressure (EIOP) with single<br>topical agent for intervention;<br>no visual field deficit | EIOP causing early visual<br>field deficits; multiple topical<br>or oral agents indicated;<br>limiting instrumental ADL | EIOP causing marked visual<br>field deficits (e.g., involving<br>both superior and inferior<br>visual fields); operative<br>intervention indicated;<br>limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |
| | cterized by an increase in pressu | 1 | i i | | |
| Keratitis | - | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Decline in vision (worse than<br>20/40 but better than<br>20/200); limiting self care<br>ADL | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | - |
| Definition: A disorder character<br>Night blindness | Symptomatic but not limiting | 1 | Limiting self care ADL | Blindness (20/200 or worse) | - |
| ragat billidiless | ADL | Laming institutional ADL | Lamining Sell Care ADL | in the affected eye | |
| | cterized by an inability to see clea | arly in dim light | | | |

| | | Eye dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only erized by involvement of the op | eye (20/40 or better) | Limiting vision in the affected eye (worse than 20/40 but better than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| | | | | Diadass (20/200 saussa) | |
| Papilledema | Asymptomatic; no visual field defects | vision; visual field defect<br>present sparing the central<br>20 degrees | Marked visual field defect<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by swelling around the o | otic disc. | | | I |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | erized by fear and avoidance of | light. | T | T | |
| Retinal detachment | Asymptomatic | Exudative and visual acuity<br>20/40 or better | Rhegmatogenous or<br>exudative detachment;<br>operative intervention<br>indicated; decline in vision<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | ·<br>erized by the separation of the i | nner retina layers from the unc | Ierlying pigment epithelium. | • | • |
| Retinal tear | - | Laser therapy or pneumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by a small laceration of t | ne retina, this occurs when the | vitreous separates from the re | tina. Symptoms include flashes | and floaters. |
| Retinal vascular disorder | - | Topical medication indicated | Intravitreal medication; operative intervention indicated | - | - |
| Definition: A disorder characte | erized by pathological retinal blo | ood vessels that adversely affe | cts vision. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked decrease in visual acuity (worse than 20/40); disabling; limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder involving | g the retina. | | | | |
| Scleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20/40 or better) | Symptomatic, limiting self<br>care ADL; marked decrease<br>in visual acuity (worse than<br>20/40) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by involvement of the scl | era of the eye. | <u> </u> | T | T |
| Uveitis | Asymptomatic; clinical or diagnostic observations only | Anterior uveitis; medical intervention indicated | Posterior or pan-uveitis | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by inflammation to the uv | rea of the eye. | | | I |
| Vitreous hemorrhage | Asymptomatic or mild symptoms; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL; vitrectomy indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder characte | erized by blood extravasation in | to the vitreous humor. | | | T |
| Watering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | - | - |
| Definition: A disorder of exces | ssive tearing in the eyes; it can | be caused by overproduction o | of tears or impaired drainage of | the tear duct. | T |
| Eye disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately sight-<br>threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Sight-threatening<br>consequences; urgent<br>intervention indicated;<br>blindness (20/200 or worse)<br>in the affected eye | - |

| | | Gastrointestinal dis | order 3 | | |
|---|---|---|---|---|---|
| | | I | Grade | T | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal distension | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by swelling of the abdomen. | T | I | <u> </u> | |
| Abdominal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | red by a sensation of marked disco | omfort in the abdominal region. | T | T | 1 |
| Anal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal communication | between the opening in the anal | canal to the perianal skin. | | |
| Anal hemorrhage Definition: A disorder characteriz | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Anal mucositis | Asymptomatic or mild | Symptomatic; medical | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| Ariai mucosius | symptoms; intervention not indicated | intervention indicated; limiting instrumental ADL | care ADL | urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by inflammation of the mucous | membrane of the anus. | T | T | |
| Anal necrosis | - | - | TPN or hospitalization indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | red by a necrotic process occurring | g in the anal region. | T | T | |
| Anal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by a sensation of marked disco | omfort in the anal region. | T | T | |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated; TPN or hospitalization<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by a narrowing of the lumen of | the anal canal. | T | T | |
| Anal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the anal ca | nal. | |
| Ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by accumulation of serous or h | emorrhagic fluid in the peritoneal | cavity. | T | |
| Bloating | No change in bowel function or oral intake | Symptomatic, decreased oral intake; change in bowel function | - | - | - |
| Definition: A disorder characterize | zed by subject-reported feeling of u | incomfortable fullness of the abdo | men. | T | |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the cecum. | | | | |
| Cheilitis | Asymptomatic; clinical or diagnostic observations only; | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | - | - |
| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Colitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe abdominal pain; change<br>in bowel habits; medical<br>intervention indicated;<br>peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the colon. | T | T | T | |
| Colonic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the large intestine and a | another organ or anatomic site. | T | 1 |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the colon. | | | T | 1 |
| Colonic obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | erized by blockage of the normal flow | | | Life the second | Daath |
| Colonic perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by a rupture in the colonic wall. | | | 1.26. (1)( | D II |
| Colonic stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the colon. | | | |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ry and necrotic erosive lesion on t | he mucosal surface of the colon. | | |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with regular use of laxatives or enemas; limiting instrumental ADL | Obstipation with manual evacuation indicated; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by irregular and infrequent or d | ifficult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis<br>or periapical abscess or<br>resulting in tooth loss | - | - |
| Definition: A disorder characte | erized by the decay of a tooth, in whice | h it becomes softened, discolored | and/or porous. | I | I |
| Diarrhea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day<br>over baseline; moderate<br>increase in ostomy output<br>compared to baseline | Increase of >=7 stools per day<br>over baseline; incontinence;<br>hospitalization indicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by frequent and watery bowel n | novements. | Г | Т | 1 |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to adequately aliment orally; tube feeding or TPN indicated; unstimulated saliva <0.1 ml/min | - | - |
| | erized by reduced salivary flow in the | ı | 1 | 1 | |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between the duodenum and ano | ther organ or anatomic site. | 1 | |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the duodenur | n. | T | 1 | |
| Duodenal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization or elective operative intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by blockage of the normal flow | of stomach contents through the | duodenum. | | |
| Duodenal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a rupture in the duodenal wa | all. | T | | |
| Duodenal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a narrowing of the lumen of | the duodenum. | | | |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a circumscribed, inflammato | | | nal wall.<br>T | |
| Dyspepsia | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | rized by an uncomfortable, often pai | nful feeling in the stomach, resulting | ng from impaired digestion. Sympt | oms include burning stomach, blo | ating, |
| heartburn, nausea and vomitin | | | | | <b>.</b> |
| Dysphagia | Symptomatic, able to eat regular diet | Symptomatic and altered eating/swallowing | Severely altered<br>eating/swallowing; tube feeding<br>or TPN or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by difficulty in swallowing. | | | | |
| Enterocolitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe or persistent abdominal pain; fever; ileus; peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by inflammation of the small ar | nd large intestines. | _ | , | |
| Enterovesical fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; noninvasive intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between the urinary bladder and | the intestine. | | |
| Esophageal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between the esophagus and and | ther organ or anatomic site. | • | |
| Esophageal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the esophagu | is. | | | |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Esophageal necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| efinition: A disorder characteri | zed by a necrotic process occurring | g in the esophageal wall. | | | |
| Esophageal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by blockage of the normal flow | of the contents in the esophagus | | T | |
| Esophageal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the esophageal region. | | | |
| Esophageal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a rupture in the wall of the e | esophagus. | | | |
| Esophageal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a narrowing of the lumen of | the esophagus. | | | |
| Esophageal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the esopha | geal wall. | |
| Esophageal varices<br>hemorrhage | - | Self-limited; intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from esophageal v | varices. | | T | |
| Esophagitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered eating/swallowing; oral supplements indicated | Severely altered eating/swallowing; tube feeding, TPN or hospitalization indicated | | Death |
| | zed by inflammation of the esopha | | | | |
| ecal incontinence | Occasional use of pads required | | Severe symptoms; elective operative intervention indicated | - | - |
| | zed by inability to control the escap | | | | |
| Flatulence | Mild symptoms; intervention not indicated | Moderate; persistent; psychosocial sequelae | - | - | - |
| | zed by a state of excessive gas in t | | | | |
| Gastric fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest; tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between the stomach and anoth | er organ or anatomic site. | | |
| Gastric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the gastric wa | all. | | | |
| Gastric necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | T |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by a rupture in the stomach wa | II. | 1 | 1 | 1 |
| Gastric stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the stomach. | | | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; medical intervention indicated; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | red by a circumscribed, inflammato | | | | 5 " |
| Gastritis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; medical intervention indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the stomach | | Ι | I | |
| Gastroesophageal reflux disease | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | ted by reflux of the gastric and/or d<br>result in injury to the esophageal m | | · - | nd usually caused by incompetend | e of the lowe |
| Gastrointestinal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between any part of the gastroin | testinal system and another organ | or anatomic site. | 1 |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the gastrointestinal region | 1. | T | 1 |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to maintain nutrition with dietary and lifestyle modifications; may need pharmacologic intervention | Weight loss; refractory to medical intervention; unable to maintain nutrition orally | - | - |
| Definition: A disorder characteriz | ed by an incomplete paralysis of the | ne muscles of the stomach wall re | sulting in delayed emptying of the | gastric contents into the small inte | estine. |
| Gingival pain | Mild pain | Moderate pain interfering with oral intake | Severe pain; inability to aliment orally | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the gingival region. | | | |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by bleeding from the hemorrho | ids. | Ι | Ι | |
| Hemorrhoids | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characteriz | ed by the presence of dilated vein | s in the rectum and surrounding a | rea. | | |
| lleal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an abnormal communication | between the ileum and another o | organ or anatomic site. | T | I |
| lleal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ted by bleeding from the ileal wall. | | | | |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| eal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of the intestinal contents in the il | leum. | 1 | |
| leal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a rupture in the ileal wall. | | | | |
| leal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the ileum. | | | |
| lleal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammate | ory and necrotic erosive lesion or | the mucosal surface of the ileum. | _ | |
| leus | | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by failure of the ileum to transp | | To a Color of the Color | 126. 0 | D 11 |
| ntra-abdominal hemorrhage | - | Medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding in the abdominal o | avity. | | | |
| Jejunal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communicatio | n between the jejunum and anoth | ner organ or anatomic site. | ' | Į. |
| Jejunal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the jejunal wa | 1 | | ' | Į. |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of the intestinal contents in the j | ejunum. | | |
| Jejunal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a rupture in the jejunal wall. | | | | |
| Jejunal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the jejunum. | | | |
| Jejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammate | ory and necrotic erosive lesion or | the mucosal surface of the jejunun | n | |
| _ip pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |

| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| | | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Lower gastrointestinal<br>hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the lower gas | trointestinal tract (small intestine, | large intestine, and anus). | | |
| Malabsorption | - | Altered diet; oral intervention indicated | Inability to aliment adequately;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by inadequate absorption of nu | trients in the small intestine. Sym | ptoms include abdominal marked o | 1 | |
| Mucositis oral | Asymptomatic or mild symptoms; intervention not indicated | Moderate pain; not interfering with oral intake; modified diet indicated | Severe pain; interfering with oral intake | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by inflammation of the oral mu | cosal. | 1 | Ι | |
| Nausea | Loss of appetite without alteration in eating habits | Oral intake decreased without significant weight loss, dehydration or malnutrition | Inadequate oral caloric or fluid intake; tube feeding, TPN, or hospitalization indicated | - | - |
| | zed by a queasy sensation and/or t | | 11 | 126. (1) | D # |
| Obstruction gastric | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | zed by blockage of the normal flow | | | <u> </u> | |
| Oral cavity fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between the oral cavity and ano | ther organ or anatomic site. | | |
| Oral dysesthesia | Mild discomfort; not interfering with oral intake | Moderate pain; interfering with oral intake | Disabling pain; tube feeding or TPN indicated | - | - |
| | zed by a burning or tingling sensati | | | | |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the mouth. | | 1 | T | |
| Oral pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | | | Γ | |
| Pancreatic duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a narrowing of the lumen of | the pancreatic duct. | • | • | , |
| Pancreatic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between the pancreas and anoth | ner organ or anatomic site. | T | |
| Pancreatic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the pancreas | | | | |
| Pancreatic necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | g in the pancreas. | , | | 1 |
| Pancreatitis | - | Enzyme elevation or radiologic findings only | Severe pain; vomiting; medical intervention indicated (e.g., analgesia, nutritional support) | Life-threatening consequences; urgent intervention indicated | Death |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| efinition: A disorder characteriz | ed by inflammation of the pancrea | S. | | | |
| Periodontal disease | Gingival recession or gingivitis;<br>limited bleeding on probing; mild<br>local bone loss | Moderate gingival recession or<br>gingivitis; multiple sites of<br>bleeding on probing; moderate<br>bone loss | Spontaneous bleeding; severe bone loss with or without tooth loss; osteonecrosis of maxilla or mandible | - | - |
| efinition: A disorder in the ging | val tissue around the teeth. | | | | |
| eritoneal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | red by a necrotic process occurring | in the peritoneum. | 1 | T | |
| Proctitis | Rectal discomfort, intervention not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteriz | ed by inflammation of the rectum. | | | | |
| Rectal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the rectum and another | organ or anatomic site. | | |
| Rectal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the rectal wall | and discharged from the anus. | | | |
| Rectal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation of the mucous | membrane of the rectum. | 1 | | 1 |
| Rectal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the rectal wall. | | | |
| Rectal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by blockage of the normal flow | of the intestinal contents in the re | ctum. | 1 | 1 |
| Rectal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | red by a sensation of marked disco | _ | 0 | 126. (1 | D ! |
| ectal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| efinition: A disorder characteriz | ed by a rupture in the rectal wall. | | | | |
| dectal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| efinition: A disorder characteriz | ed by a narrowing of the lumen of | the rectum. | | | |
| lectal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function (e.g. altered dietary habits, vomiting, diarrhea) | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | i . | İ | 1 | İ | l |

| Self-imited: trianvention indicated control of the decision indicated cont | Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|---|
| Recopertoneal hemorrhage - Self-Imited: intervention inclosited of self-Imited intervention inclosited of self-Imited intervention inclosited or self-Imited intervention inclosited or self-Imited intervention inclosited or self-Imited intervention inclosited or self-Imited intervention inclosited or self-Imited intervention inclosited inter | | | | | | |
| Definition: A disorder characterized by bleeding from the retroperionneal area. Sulvary duct inflammation Slightly bleeding from the retroperionneal area. Sulvary duct inflammation Slightly bleeding from the retroperionneal area. Sulvary duct inflammation Slightly bleeding from the retroperionneal area. Acute salivary gland necrose; were secretic-induced symptoms; cap, thick salivatoral secretion-induced symptoms; cap, thick salivatoral secretion-induced symptoms; cap, thick salivatoral secretion or devices or againging in get area ADL; disabiling or Part indicated; cap part intervention indicated; cap part intervention indicated; cap part intervention indicated; cap part intervention indicated; cap part intervention and indicated or diagnostic observations only; intervention not indicated or | Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Salivary duct inflammation Slightly thickened salivis; alightly Takes replaced to the salivis district of the first control of diagnosis coherentation only, intervention of the first control of diagnosis coherentations only, intervention of the first control of diagnosis coherentations only, intervention of the first control of diagnosis coherentations only, intervention of the mucous membrane of the small intestinal obstruction Definition: A disorder characterized by inflammation of the mucous membrane of the small intestinal obstruction Abymptomatic; clinical or diagnosis coherentations only, intervention only inflammation of the mucous membrane of the small intestinal obstruction Poefinition: A disorder characterized by blockage of the normal flow of the intestinal control only intervention only inflammation of the mucous membrane of the small intestinal perforation Abuse of the first control of diagnosis coherentations only, intervention only inflammation of the mucous membrane of the small intestinal control of diagnosis coherentations only, intervention and flow of the intestinal control of diagnosis coherentations only, intervention and indicated introvention indicated introventio | · | | indicated | endoscopic, or elective | 1 | Death |
| attended in the indicated; services acception-induced symptoms; increased in the indicated; services acception or gagging); tube formation of the salvary duct. Salvary gland fietula Asymptomatic, clinical or diagnostic observations only; intervention on indicated intervention indicated intervention | | T . | | A cute adjugate aland pagagia | Life threatening concessions | Dooth |
| degnostic observations only; intervention indicated intervention indicated intervention indicated symptoms; intervention not indicated intervention indicated; limiting self-care ADL. Definition: A disorder characterized by inflammation of the mucus membrane of the small intestine. Small intestinal obstruction | Salivary duct inflammation | 1 | markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms; | severe secretion-induced<br>symptoms (e.g., thick saliva/oral<br>secretions or gagging); tube<br>feeding or TPN indicated; | _ : | Death |
| diagnostic observations only; intervention not indicated intervention not indicated of intervention not indicated of intervention indicated indicated and indicated indicated and indicated indicated indicated and indicated indicated and symptoms; intervention not indicated intervention indicated intervention indicated intervention indicated intervention indicated. Small intestinal mucositis and anymptoms; intervention not indicated intervention indicated; limiting self-care ADL indicated intervention indicated; limiting self-care ADL indicated intervention indicated; limiting self-care ADL indicated intervention indicated intervention indicated; limiting self-care ADL indicated intervention indicated interventi | Definition: A disorder characteriz | zed by inflammation of the salivary | duct. | | | |
| Small intestinal mucositis Asymptomatic or mild symptoms; intervention not indicated; mining instrumental ADL intervention indicated; limiting self care ADL. Definition: A disorder characterized by inflammation of the mucous membrane of the small intestinal obstruction Agymptomatic; clinical or diagnostic observations only; intervention indicated with real additional and appropriate intervention indicated with real and appro | Salivary gland fistula | diagnostic observations only; | | hospitalization indicated; elective operative intervention | urgent operative intervention | Death |
| symptoms, intervention not indicated, imiting instrumental ADL self-care ADL indicated with indicated indicated, imiting self-care ADL self-care ADL symptomatic, clinical or diagnostic observations only, intervention not indicated intervention indicated by blockage of the normal flow of the intestinal contents. Small intestinal perforation Definition: A disorder characterized by blockage of the normal flow of the intestinal contents. Small intestinal perforation Definition: A disorder characterized by a care and intervention indicated Definition: A disorder characterized by a care and intervention indicated intervention indicated Definition: A disorder characterized by a number of the small intestine wall. Small intestinal stenosis Asymptomatic, clinical or diagnostic observations only, intervention not indicated Definition: A disorder characterized by a narrowing of the lumen of the small intestine. Small intestine ulcer Asymptomatic, clinical or diagnostic observations only, intervention indicated Definition: A disorder characterized by a narrowing of the lumen of the small intestine. Small intestine ulcer Asymptomatic, clinical or diagnostic observations only, intervention indicated Definition: A disorder characterized by a circumscribed, inflammatory and necrotic crosive lesion on the mucosal surface of the small intestine. Stomach pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL; disabling Severe pain; limiting self care ADL; disabling Severe pain; limiting self care ADL; disabling Definition: A disorder characterized by a sensation of marked discomflot in the stomach. Tooth development disorder Asymptomatic; planead of the small intestine. Insurance ADL In | Definition: A disorder characteriz | zed by an abnormal communication | between a salivary gland and an | other organ or anatomic site. | | |
| Small intestinal obstruction diagnostic cibrical or diagnostic cobservations only; intervention not indicated intervention indicated indicated; one-mergent operative intervention indicated intervention indi | Small intestinal mucositis | symptoms; intervention not | intervention indicated; limiting | intake; tube feeding, TPN or hospitalization indicated; limiting | | Death |
| diagnostic observations only; intervention not indicated with performance of the small intestinal stenosis and indicated control indicated of diagnostic observations only; intervention indicated or operative intervention indicated or poperative or endoscopic intervention indicated; ilentiting self care ADL; disabling or the sum of the su | Definition: A disorder characteriz | ed by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal perforation | Small intestinal obstruction | diagnostic observations only; | function; limiting instrumental | elective operative intervention indicated; limiting self care ADL; | urgent operative intervention | Death |
| Definition: A disorder characterized by a rupture in the small intestine wall. Small intestinal stenosis Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a narrowing of the lumen of the small intestine. Small intestine ulcer Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a narrowing of the lumen of the small intestine. Small intestine ulcer Asymptomatic; clinical or diagnostic observations only; intervention not indicated Asymptomatic; clinical or diagnostic observations only; intervention not indicated Apulation Asymptomatic; clinical or diagnostic observations only; intervention not indicated ADL Definition: A disorder characterized by a circumscribed, inflammatory and necrotic erosive lesion on the mucosal surface of the small intestine. Stomach pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by a sensation of marked discontrol tooth or enamel tooth or enamel Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth development disorder Surface stains Asymptomatic; altered GI surton, tube feeding, TPN or hospitalization indicated Symptomatic; altered GI function; tube feeding, TPN or hospitalization indicated Severely altered GI function; TPN indicated; elective operative or endoscopic intervention indicated; limiting self care ADL; disabling Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discontrol in the stomach. Tooth development disorder Asymptomatic; altered GI surton. The indicated: function; tube feeding, TPN or hospitalization indicated Symptomatic; altered GI function; TPN indicated; leactive operative intervention indicated Severe pain; limiting self care ADL | Definition: A disorder characteriz | zed by blockage of the normal flow | of the intestinal contents. | | | |
| Asymptomatic; clinical or diagnostic observations only; intervention not indicated Symptomatic; altered GI function; tube feeding, TPN or hospitalization indicated operative intervention indicated; non-emergent operative intervention indicated. Severely altered GI function; tube feeding, TPN or hospitalization indicated operative intervention indicated. Severely altered GI function; tube feeding, TPN or hospitalization indicated. Severely altered GI function; tintervention indicated. Severely altered GI function; TPN indicated; elective operative or endoscopic intervention indicated. ADL Definition: A disorder characterized by a circumscribed, inflammatory and necrotic erosive lesion on the mucosal surface of the small intestine. Stomach pain Mild pain Moderate pain; limiting instrumental ADL ADL Definition: A disorder characterized by a sensation of marked discomfort in the stomach. Tooth development disorder Asymptomatic; hypoplasia of tooth or enamel surgery Impairment correctable with oral surgery limiting tooth development. Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains | Small intestinal perforation | - | | | urgent operative intervention | Death |
| diagnostic observations only; intervention not indicated function altered GI function; tube feeding, TPN or hospitalization indicated indicated; non-emergent operative intervention indicated Definition: A disorder characterized by a narrowing of the lumen of the small intestine. Small intestine ulcer Asymptomatic; clinical or diagnostic observations only; intervention not indicated ADL Symptomatic; altered GI function; TPN indicated; elective operative or endoscopic intervention indicated; imiting self care ADL; disabling Definition: A disorder characterized by a circumscribed, inflammatory and necrotic erosive lesion on the mucosal surface of the small intestine. Stomach pain Mild pain Moderate pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the stomach. Toth development disorder Asymptomatic; hypoplasia of toth or enamel Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Toth discoloration Surface stains Definition: A disorder characterized by a change in tooth hue or tint. Toothache Mild pain Moderate pain; limiting Severe pain; limiting instrument with impairment not surgically correctable; disabling Severe pain; limiting and the surgically correctable; disabling Definition: A disorder characterized by a change in tooth hue or tint. | Definition: A disorder characterize | zed by a rupture in the small intesti | ne wall. | | | |
| Small intestine ulcer Asymptomatic; clinical or diagnostic observations only; intervention not indicated ADL Symptomatic; altered GI function; TPN indicated; elective operative or endoscopic intervention indicated; limiting self care ADL; disabling Definition: A disorder characterized by a circumscribed, inflammatory and necrotic erosive lesion on the mucosal surface of the small intestine. Stomach pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by a sensation of marked discomfort in the stomach. Tooth development disorder Asymptomatic; hypoplasia of tooth or enamel Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains Definition: A disorder characterized by a change in tooth hue or tint. Moderate pain; limiting self care ADL Maldevelopment with impairment not surgically correctable; disabling | Small intestinal stenosis | diagnostic observations only; | | altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent | urgent operative intervention | Death |
| diagnostic observations only; intervention not indicated hDL limiting instrumental ADL and necrotic erosive lesion on the mucosal surface of the small intestine. Stomach pain Mild pain Moderate pain; limiting instrumental ADL has provided in the stomach. Tooth development disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains - Definition: A disorder characterized by a change in tooth hue or tint. Midd pain Moderate pain; limiting self care ADL has provided intervention indicated; limiting self care ADL; disabling has perative or endoscopic intervention indicated; limiting self care application to the mucosal surface of the small intestine. Severe pain; limiting self care ADL has provided intervention indicated; limiting self care application to the mucosal surface of the small intestine. Severe pain; limiting self care application to the stomach. - Tooth development disorder has pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains | Definition: A disorder characteriz | zed by a narrowing of the lumen of | the small intestine. | | | |
| Stomach pain Mild pain Moderate pain; limiting instrumental ADL Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the stomach. Tooth development disorder Asymptomatic; hypoplasia of tooth or enamel surgery Impairment correctable with oral surgery correctable; disabling Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains Definition: A disorder characterized by a change in tooth hue or tint. Toothache Mild pain Moderate pain; limiting Severe pain; limiting self care | Small intestine ulcer | diagnostic observations only; | function; limiting instrumental | TPN indicated; elective operative or endoscopic intervention indicated; limiting | urgent operative intervention | Death |
| instrumental ADL Definition: A disorder characterized by a sensation of marked discomfort in the stomach. Tooth development disorder Asymptomatic; hypoplasia of tooth or enamel Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains Definition: A disorder characterized by a change in tooth hue or tint. Toothache Mild pain Moderate pain; limiting Severe pain; limiting self care ADL ADL ADL ADL ADL ADL ADL | Definition: A disorder characteriz | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on t | the mucosal surface of the small in | ntestine. | |
| Tooth development disorder Asymptomatic; hypoplasia of tooth or enamel surgery Impairment correctable with oral surgically correctable; disabling Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains | Stomach pain | Mild pain | · | _ · · · · · · · | - | - |
| tooth or enamel surgery impairment not surgically correctable; disabling Definition: A disorder characterized by a pathological process of the teeth occurring during tooth development. Tooth discoloration Surface stains Definition: A disorder characterized by a change in tooth hue or tint. Toothache Mild pain Moderate pain; limiting Severe pain; limiting self care | Definition: A disorder characterize | zed by a sensation of marked disco | omfort in the stomach. | Τ | Τ | |
| Tooth discoloration Surface stains Definition: A disorder characterized by a change in tooth hue or tint. Toothache Mild pain Moderate pain; limiting Severe pain; limiting self care | Tooth development disorder | 1 | | impairment not surgically | - | - |
| Definition: A disorder characterized by a change in tooth hue or tint. Toothache Mild pain Moderate pain; limiting Severe pain; limiting self care | Definition: A disorder characterize | red by a pathological process of the | e teeth occurring during tooth deve | elopment. | Т | |
| Toothache Mild pain Moderate pain; limiting Severe pain; limiting self care | Tooth discoloration | Surface stains | - | - | - | - |
| | Definition: A disorder characterize | zed by a change in tooth hue or tin | i. | 1 | 1 | |
| | Toothache | Mild pain | | _ · · · · · · · | - | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Typhlitis | - | - | Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritoneal signs | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the cecum. | ' | | ' | 1 |
| Upper gastrointestinal<br>hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | zed by bleeding from the upper gas | strointestinal tract (oral cavity, pha | rynx, esophagus, and stomach). | | |
| Vomiting | 1 - 2 episodes (separated by 5 minutes) in 24 hrs | 3 - 5 episodes (separated by 5 minutes) in 24 hrs | >=6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | zed by the reflexive act of ejecting | the contents of the stomach through | gh the mouth. | | |
| Gastrointestinal disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | disabling; limiting self care ADL | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Chills | Mild sensation of cold;<br>shivering; chattering of teeth | Moderate tremor of the entire body; narcotics indicated | Severe or prolonged, not responsive to narcotics | - | - |
| Definition: A disorder charact | erized by a sensation of cold that ofter | n marks a physiologic response to | sweating after a fever. | | |
| Death neonatal | - | - | - | - | Death |
| Definition: A disorder charact | erized by cessation of life occurring du | uring the first 28 days of life. | • | | , |
| Death NOS | - | - | - | - | Death |
| Definition: A cessation of life | that cannot be attributed to a CTCAE | term associated with Grade 5. | ' | • | |
| Edema face | Localized facial edema | Moderate localized facial edema; limiting instrumental ADL | Severe swelling; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by swelling due to excessive flu | uid accumulation in facial tissues. | 1 | 1 | |
| Edema limbs | 5 - 10% inter-limb discrepancy in volume or circumference at point of greatest visible difference; swelling or obscuration of anatomic architecture on close inspection | >10 - 30% inter-limb<br>discrepancy in volume or<br>circumference at point of<br>greatest visible difference;<br>readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | >30% inter-limb discrepancy in<br>volume; gross deviation from<br>normal anatomic contour;<br>limiting self care ADL | - | - |
| Definition: A disorder charact | erized by swelling due to excessive flu | ı<br>ıid accumulation in the upper or lo | wer extremities. | 1 | 1 |
| Edema trunk | Swelling or obscuration of anatomic architecture on close inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | Gross deviation from normal anatomic contour; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by swelling due to excessive flu | ! | I | 1 | 1 |
| Facial pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Definition: A disorder charact | erized by a sensation of marked disco | omfort in the face. | ! | 1 | 1 |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest;<br>limiting instrumental ADL | Fatigue not relieved by rest, limiting self care ADL | - | - |
| Definition: A disorder charact | erized by a state of generalized weak | | | omplish daily activities. | |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) | >40.0 degrees C (>104.0 degrees F) for <=24 hrs | >40.0 degrees C (>104.0 degrees F) for >24 hrs | Death |
| Definition: A disorder charact | erized by elevation of the body's temp | erature above the upper limit of n | ormal. | 1 | |
| Flu like symptoms | Mild flu-like symptoms present | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | | - |
| cough. | erized by a group of symptoms similar | to those observed in patients with | it the na. It includes level, chills, b | ody acries, maiaise, ioss or appeti | ie and di |
| Gait disturbance | Mild change in gait (e.g., wide-<br>based, limping or hobbling) | Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental ADL | Disabling; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by walking difficulties | I | I | 1 | I |
| Hypothermia | - | 35 - >32 degrees C; 95 - >89.6 degrees F | 32 - >28 degrees C; 89.6 -<br>>82.4 degrees F | <=28 degrees C; 82.4 degrees<br>F; life-threatening<br>consequences (e.g., coma,<br>hypotension, pulmonary edema,<br>acidemia, ventricular fibrillation) | Death |

| General disorders and administration site conditions | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Infusion related reaction | Mild transient reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic | | Life-threatening consequences; urgent intervention indicated | Death |
| | | medications indicated for <=24 hrs | following initial improvement; hospitalization indicated for clinical sequelae | | |
| | zed by adverse reaction to the infus | | | | - · |
| Infusion site extravasation | - | Erythema with associated symptoms (e.g., edema, pain, induration, phlebitis) | Ulceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by leakage of a pharmacologic sation and marked discomfort at the | = | nfusion site into the surrounding ti | ssue. Signs and symptoms include | e induration, |
| Injection site reaction | Tenderness with or without associated symptoms (e.g., warmth, erythema, itching) | Pain; lipodystrophy; edema; phlebitis | Ulceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an intense adverse reaction | (usually immunologic) developing | at the site of an injection. | T | |
| Irritability | Mild; easily consolable | Moderate; limiting instrumental ADL; increased attention indicated | Severe abnormal or excessive response; limiting self care ADL; inconsolable | - | - |
| Definition: A disorder characteri condition. | zed by an abnormal responsivenes | s to stimuli or physiological arousa | al; may be in response to pain, frig | ht, a drug, an emotional situation o | or a medical |
| Localized edema | Localized to dependent areas, | Moderate localized edema and | Severe localized edema and | - | - |
| | no disability or functional impairment | intervention indicated; limiting instrumental ADL | intervention indicated; limiting self care ADL | | |
| Definition: A disorder characteri | zed by swelling due to excessive flu | uid accumulation at a specific ana | tomic site. | ' | ı |
| Malaise | Uneasiness or lack of well being | Uneasiness or lack of well being; limiting instrumental ADL | - | - | - |
| Definition: A disorder characteri | uzed by a feeling of general discomf | | feeling. | ı | ı |
| Multi-organ failure | - | - | Shock with azotemia and acid- | Life-threatening consequences | Death |
| · · | | | base disturbances; significant coagulation abnormalities | (e.g., vasopressor dependent<br>and oliguric or anuric or<br>ischemic colitis or lactic<br>acidosis) | |
| Definition: A disorder characteri | zed by progressive deterioration of | the lungs, liver, kidney and clotting | g mechanisms. | | |
| Neck edema | Asymptomatic localized neck edema | Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL | Generalized neck edema (e.g., difficulty in turning neck); limiting self care ADL | - | - |
| Definition: A disorder characteri | l<br>zed by swelling due to an accumula | ı | I | I | l |
| Non-cardiac chest pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Definition: A disorder characteri | I<br>zed by discomfort in the chest unre | ı | MUL | I | |
| Pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | l<br>zed by the sensation of marked dis | ı | ADL | | |
| Sudden death NOS | - | - | _ | _ | Death |
| | -<br>ation of life that cannot be attributed | I to a CTCΔF term associated with | Grade 5 | I | Death |
| General disorders and | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life threatening concessioness: | Death |
| deficient disorders and administration site conditions - Other, specify | symptomatic of fillid<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | noninvasive intervention indicated; limiting age-appropriate instrumental ADL | but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing | Life-threatening consequences; urgent intervention indicated | Dealli |
| | | | hospitalization indicated;<br>disabling; limiting self care ADL | | |

| | | Hepatobiliary diso | rders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bile duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; IV fluids indicated <24<br>hrs | Severely altered GI function;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the bile duct. | 1 | ı | 1 |
| Biliary fistula | - | Symptomatic and intervention not indicated | Severely altered GI function;<br>TPN indicated; endoscopic<br>intervention indicated; elective<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the bile ducts and anoth | ner organ or anatomic site. | | 1 |
| Cholecystitis | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the g | allbladder. It may be associated w | vith the presence of gallstones. | | |
| Gallbladder fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Symptomatic or severely altered<br>GI function; TPN indicated;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | n between the gallbladder and and | ther organ or anatomic site. | Т | 1 |
| Gallbladder necrosis | - | - | - | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the gallbladder. | | | |
| Gallbladder obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; IV fluids indicated <24<br>hrs | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by blockage of the normal flow | of the contents of the gallbladder. | T | | |
| Gallbladder pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the gallbladder region. | T | Γ | 1 |
| Gallbladder perforation | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the gallbladder | wall. | | | 1 |
| Hepatic failure | - | - | Asterixis; mild encephalopathy; limiting self care ADL | Moderate to severe encephalopathy; coma; life-threatening consequences | Death |
| | | etabolize chemicals in the body. La | aboratory test results reveal abnor | mal plasma levels of ammonia, bi | lirubin, lactic |
| dehydrogenase, and alkaline pho | 1 | O | Towns for the Control of | I if the state of | Death |
| Hepatic hemorrhage | Mild; intervention not indicated | Symptomatic; medical intervention indicated | Transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the liver. | | | | |
| Hepatic necrosis | - | - | - | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the hepatic parenchyma. | 1 | ı | |
| Hepatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by a sensation of marked disco | omfort in the liver region. | T | <b>.</b> | |
| Perforation bile duct | - | - | Radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the wall of the e | xtrahepatic or intrahepatic bile due | ct. | | |

| | | Hepatobiliary diso | rders | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Portal hypertension | - | Decreased portal vein flow | Reversal/retrograde portal vein flow; associated with varices and/or ascites | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an increase in blood pressu | re in the portal venous system. | | | |
| Portal vein thrombosis | - | Intervention not indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by the formation of a thrombus | (blood clot) in the portal vein. | | | |
| Hepatobiliary disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | disabling; limiting self care ADL | | |

| | | Immune system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Allergic reaction | Transient flushing or rash, drug<br>fever <38 degrees C (<100.4<br>degrees F); intervention not<br>indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an adverse local or general | response from exposure to an alle | ergen.<br>T | T | |
| Anaphylaxis | - | - | Symptomatic bronchospasm,<br>with or without urticaria;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an acute inflammatory react resents with breathing difficulty, dia | <del>-</del> | | <del>-</del> | ypersensitivity |
| Autoimmune disorder | Asymptomatic; serologic or other evidence of autoimmune reaction, with normal organ function; intervention not indicated | Evidence of autoimmune reaction involving a non-essential organ or function (e.g., hypothyroidism) | Autoimmune reactions involving major organ (e.g., colitis, anemia, myocarditis, kidney) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder resulting fro | om loss of function or tissue destru | iction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses of the individe | ual to his own |
| Cytokine release syndrome | Mild reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| Definition: A disorder characteriz | ed by nausea, headache, tachycai | rdia, hypotension, rash, and short | ness of breath; it is caused by the | release of cytokines from the cells | i |
| Serum sickness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate arthralgia; fever, rash, urticaria, antihistamines indicated | extensive rash; steroids or IV fluids indicated | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| | ed by a delayed-type hypersensitive foreign antigen. Symptoms include | = : | | | = |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| | zed by an infectious process involv | | n | I | <b>5</b> " |
| Anorectal infection | Localized; local intervention | Oral intervention indicated (e.g., | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | indicated | antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic, endoscopic, or | urgent intervention indicated | |
| | | | operative intervention indicated | | |
| Definition: A disorder character | l<br>zed by an infectious process involv | ing the anal area and the rectum | operative intervention indicated | l | |
| Appendicitis | zed by all illections process illvolv | ing the arial area and the rectum. | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| френцісніѕ | - | _ | antiviral intervention indicated; | urgent intervention indicated | Dealii |
| | | | radiologic or operative | digent intervention indicated | |
| | | | intervention indicated | | |
| Nafinikian. A dinandan abanaskan | | | • | | |
| | zed by acute inflammation to the ve | | | l ife there are in a constant | Daath |
| Appendicitis perforated | - | Symptomatic; medical | Severe symptoms; elective | Life-threatening consequences; | Death |
| Daginialana Andrewski i i i i | and hor and a transfer of the second | intervention indicated | operative intervention indicated | urgent intervention indicated | |
| | zed by acute inflammation to the vertile eal wall rupture causes the release | | | | ıne |
| Arteritis infective | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | 23411 |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing an artery. | • | 1 | ' |
| Biliary tract infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| • | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the biliary tract. | | | |
| Bladder infection | - | Oral intervention indicated (e.g., | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | antibiotic, antifungal, antiviral) | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic, endoscopic, or | | |
| | | | operative intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the bladder. | | 1 | |
| Bone infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | | T | Ī | 1 |
| Breast infection | - | Local infection with moderate | Severe infection; axillary | Life-threatening consequences; | Death |
| | | symptoms; oral intervention | adenitis; IV antibacterial, | urgent intervention indicated | |
| | | indicated (e.g., antibiotic, | antifungal, or antiviral | | |
| | | antifungal, antiviral) | intervention indicated | | |
| | zed by an infectious process involv | | | | |
| Bronchial infection | - | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., | antiviral intervention indicated; | urgent intervention indicated | |
| | | antibiotic, antifungal, antiviral) | radiologic, endoscopic, or | | |
| Dofinition: A disease of the control | and by an infa-ti | ing the branch: | operative intervention indicated | l | l |
| | zed by an infectious process involv | | N/ (PL - P | Life the control | D |
| Catheter related infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated; oral intervention | antiviral intervention indicated; | urgent intervention indicated | |
| | | indicated (e.g., antibiotic, antifungal, antiviral) | radiologic or operative intervention indicated | | |
| | <br>zed by an infectious process that a | | Intervention mulcated | I | l |
| )efinition: Δ disorder characteri | zou by an infectious process tilat a | noco occontrary to catheter use. | IV antibiatio antifungal or | Life-threatening consequences; | Death |
| | | | | | Dealli |
| | - | - | IV antibiotic, antifungal, or | = : | |
| Definition: A disorder characteri<br>Cecal infection | - | - | antiviral intervention indicated; | urgent intervention indicated | |
| | - | - | <u> </u> | = : | |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | d by an infectious process ir | volving the cecum. | ı | 1 | |
| Cervicitis infection Definition: A disorder characterize | d by an infectious process in | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | d by an injectious process in | | NA - Children - Cf 1 | 126. 0 | D |
| Conjunctivitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | nvolving the conjunctiva. Clinical manifo | estations include pink or red color | in the eyes. | |
| Corneal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | nvolving the cornea. | | 1 | 1 |
| Cranial nerve infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | nvolving a cranial nerve. | 1 | 1 | |
| Device related infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | nvolving the use of a medical device. | | 1 | 1 |
| Duodenal infection | - | Moderate symptoms; medical intervention indicated (e.g., oral antibiotics) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | volving the duodenum. | | | |
| Encephalitis infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>severe changes in mental<br>status; self-limited seizure<br>activity; focal neurologic<br>abnormalities | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | volving the brain tissue. | | | |
| Encephalomyelitis infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | nvolving the brain and spinal cord tissu | es. | | |
| Endocarditis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | d by an infectious process ir | nvolving the endocardial layer of the he | eart. | | |
| Endophthalmitis | - | Local intervention indicated | Systemic intervention or | Blindness (20/200 or worse) | - |

| per 24 hrs or duration of illness 248 hrs; moderate abdominal pain antiviral inter adiologic, er operative interprofuse wate signs of hypo diarrhes. Esophageal infection Definition: A disorder characterized by an infectious process involving the small and large intestines. Esophageal infection - Local intervention indicated (e.g., oral antibiotic, antifungal, antiviral) indicated indicated indicated (e.g., oral antibiotic, antifungal, antiviral intervention indicated (e.g., topical antibiotic, antifurial intervention indicated (e.g., topical antibiotic, antifurial intervention indicated (e.g., topical antibiotic, antifurial intervention indicated (e.g., topical antibiotic, antifurial intervention indicated intervention ind | antifungal, or vention indicated; operative indicated antifungal, or vention indicated urgent intervention indicated antifungal, or vention indicated; operative Life-threatening consequence urgent intervention indicated; operative | s; Death |
|---|---|---|
| Interocolitis infectious - Passage of >3 unformed stools per 24 hrs or duration of illness >48 hrs; moderate abdominal pain Definition: A disorder characterized by an infectious process involving the small and large intestines. Esophageal infection - Local intervention indicated (e.g., oral antibiotic, antifungal, antiviral) Definition: A disorder characterized by an infectious process involving the esophagus. Esperintion: A disorder characterized by an infectious process involving the esophagus. Definition: A disorder characterized by an infectious process involving the esophagus. Esperintion: A disorder characterized by an infectious process involving the esophagus. Definition: A disorder characterized by an infectious process involving the esophagus. Definition: A disorder characterized by an infectious process involving the esophagus. Definition: A disorder characterized by an infectious process involving the eye. Salibladder infection - Vanitibiotic, antifungal, or antiviral) IV antibiotic, antiviral inter radiologic, or operative intervention indicated (e.g., antibiotic) antiviral inter radiologic, or operative intervention indicated (e.g., antibiotic) antiviral inter radiologic, or operative intervention indicated (e.g., antibiotic) antiviral inter radiologic, or operative intervention indicated (e.g., antibiotic, antiviral) Definition: A disorder characterized by an infectious process involving the gums. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by an infectious process involving the liver parenchyma. Definition: A disorder characterized by an infectious process involving the liv | antifungal, or vention indicated; andoscopic, or ervention indicated; ary diarrhea with evolemia; bloody er; severe ain; hospitalization antifungal, or vention indicated; operative indicated antifungal, or vention indicated; operative indicated; operative operative enucleation Life-threatening consequence urgent intervention indicated; or urgent intervention indicated; enucleation | s; Death |
| per 24 hrs or duration of illness antiviral inter radiologic, er operative interprofuse wate signs of hypo diarrhes. Sophageal infection Definition: A disorder characterized by an infectious process involving the small and large intestines. Sophageal infection - Local intervention indicated (e.g., oral antibiotic, antifungal, antiviral) Definition: A disorder characterized by an infectious process involving the esophagus. Vey infection - Localized: local intervention indicated (e.g., topical antibiotic, antifural) Definition: A disorder characterized by an infectious process involving the eye. Definition: A disorder characterized by an infectious process involving the eye. Definition: A disorder characterized by an infectious process involving the gallbladder. Soun infection - Vanitibiotic, antifungal, or antiviral inter radiologic, or operative into indicated (e.g., antibiotic, antifungal, antiviral) Definition: A disorder characterized by an infectious process involving the gallbladder. Soun infection Local therapy indicated (swish and swallow) Definition: A disorder characterized by an infectious process involving the gallbladder. Definition: A disorder characterized by an infectious process involving the gams. Hepatic infection - Vanitibiotic, antifungal, antiviral) Definition: A disorder characterized by an infectious process involving the gams. Hepatic infection - Vanitibiotic, antifungal, antiviral inter radiologic or intervention indicated (e.g., topical antibiotic, antiviral inter radiologic or intervention indicated (e.g., topical antibiotic, antiviral inter radiologic or intervention indicated (e.g., topical antibiotic, antiviral inter radiologic or intervention indicated (e.g., topical antibiotic, antiviral) Definition: A disorder characterized by an infectious process involving the liver. | vention indicated; andoscopic, or ervention indicated; ary diarrhea with poolemia; bloody er; severe ain; hospitalization antifungal, or vention indicated; operative indicated antifungal, or vention indicated; operative indicated antifungal, or vention indicated; operative indicated; operative indicated; operative indicated; operative | s; Death |
| Definition: A disorder characterized by an infectious process involving the small and large intestines. Esophageal infection - Local intervention indicated (e.g., oral antibiotic, antifungal, antiviral) IV antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic, erroperative intervention indicated (e.g., antibiotic, antiviral interradiologic, erroperative intervention indicated (e.g., antibiotic, antiviral) Definition: A disorder characterized by an infectious process involving the gallbladder. Gaum infection Local therapy indicated (swish and swallow) Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) Poefinition: A disorder characterized by an infectious process involving the gums. Hepatic infection Definition: A disorder characterized by an infectious process involving the liver. Hepatic infection Asymptomatic, treatment not indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Poefinition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Poefinition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Localized, local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) IV antibiotic, antifungal, or antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | rvention indicated; operative indicated antifungal, or rvention indicated; operative urgent intervention indicated; operative urgent intervention indicated; operative | s; Death |
| Local intervention indicated (e.g., oral antibiotic, antifungal, antiviral interradiologic or intervention indicated (e.g., oral antibiotic, antifungal, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) IV antibiotic, antifungal, or antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) IV antibiotic, antifungal, or antiviral) IV antibiotic, antifungal, or antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated intervention indicated (e.g., antibiotic, antiviral interradiologic, eroperative intervention indicated (e.g., antibiotic, antifungal, antiviral) IV antibiotic, antiviral interradiologic or intervention indicated (e.g., antibiotic, antiviral) IV antibiotic, antiviral interradiologic or intervention indicated (e.g., antibiotic, antiviral) IV antibiotic, antiviral interradiologic or intervention indicated (e.g., antiviral interradiologic or intervention indicated (e.g., antiviral) IV antibiotic, a | rvention indicated; operative indicated antifungal, or rvention indicated; operative urgent intervention indicated; operative urgent intervention indicated; operative | s; Death |
| (e.g., oral antibiotic, antifungal, antiviral interradiologic or intervention i Definition: A disorder characterized by an infectious process involving the esophagus. | rvention indicated; operative indicated antifungal, or rvention indicated; operative urgent intervention indicated; operative urgent intervention indicated; operative | s; Death |
| Localized; local intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral) Definition: A disorder characterized by an infectious process involving the eye. Sum infection Local therapy indicated (swish and swallow) Definition: A disorder characterized by an infectious process involving the gallbladder. Sum infection Local therapy indicated (swish and swallow) Definition: A disorder characterized by an infectious process involving the gallbladder. Sum infection Local therapy indicated (swish and swallow) Definition: A disorder characterized by an infectious process involving the gallbladder. Sum infection Local therapy indicated (swish and swallow) Definition: A disorder characterized by an infectious process involving the gums. Hepatic infection - Definition: A disorder characterized by an infectious process involving the liver. Hepatitis viral Asymptomatic, treatment not indicated Asymptomatic, treatment not indicated Symptomatic fibrosis by bic cirrhosis; rea hepatitis Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Localized; local intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention interv | vention indicated; operative urgent intervention indicated; enucleation | |
| indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by an infectious process involving the eye. Sallbladder infection - | vention indicated; operative urgent intervention indicated; enucleation | |
| Gallbladder infection - | | s; Death |
| Definition: A disorder characterized by an infectious process involving the gallbladder. Gum infection Local therapy indicated (swish and swallow) Definition: A disorder characterized by an infectious process involving the gums. Definition: A disorder characterized by an infectious process involving the gums. Definition: A disorder characterized by an infectious process involving the gums. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by an infectious process involving the liver. Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Localized; local intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention indicated (e.g., topical antibiotic, antiviral interradiologic or intervention i | | s; Death |
| Local therapy indicated (swish and swallow) Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) IV antibiotic, antiviral interradiologic or intervention i | antifungal, or vention indicated; urgent intervention indicated urgent intervention indicated | |
| and swallow) intervention indicated (e.g., antiviral) antiviral intervention indicated (e.g., antiviral) antiviral intervention interve | | |
| Definition: A disorder characterized by an infectious process involving the liver. Hepatitis viral Asymptomatic, treatment not indicated Symptomatic, treatment not indicated Fibrosis by bic cirrhosis; real hepatitis Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Infective myositis - Localized; local intervention indicated (e.g., topical antibiotic, antiviral interradiologic or | | s; Death |
| Definition: A disorder characterized by an infectious process involving the liver. Hepatitis viral Asymptomatic, treatment not indicated Asymptomatic, treatment not indicated Symptomatic fibrosis by bic cirrhosis; real hepatitis Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Infective myositis - Localized; local intervention indicated (e.g., topical antibiotic, antiviral) IV antibiotic, antiviral interradiologic or intervention | • | , |
| Hepatitis viral Asymptomatic, treatment not indicated Asymptomatic, treatment not indicated Symptomatic fibrosis by bic cirrhosis; real hepatitis Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Localized; local intervention indicated (e.g., topical antibiotic, antiviral intervadiologic or intervention interventi | | s; Death |
| indicated fibrosis by bic cirrhosis; real hepatitis Definition: A disorder characterized by a viral pathologic process involving the liver parenchyma. Localized; local intervention indicated (e.g., topical antibiotic, antiviral) IV antibiotic, antiviral intervation intervention intervent | | |
| Infective myositis - Localized; local intervention indicated (e.g., topical antibiotic, antiviral interval interval interval intervention indicated (e.g., topical antibiotic, antiviral intervention intervention indicated (e.g., topical antibiotic, antiviral intervention interv | c liver dysfunction; opsy; compensated (e.g., ascites, coagulopathy, encephalopathy, coma) | Death |
| indicated (e.g., topical antibiotic, antiviral inter antifungal, or antiviral) radiologic or intervention i | | |
| Definition: A disorder characterized by an infectious process involving the skeletal muscles | vention indicated; operative urgent intervention indicated | s; Death |
| Sommitten. A disorder dilaracterized by an infectious process involving the skeletal inuscies. | | |
| | | s; Death |
| Definition: A disorder characterized by an infectious process involving a joint. | intervention g., drainage) or e.g., open surgical | 1 |
| Kidney infection - IV antibiotic, antiviral inter radiologic, er operative inte | g., drainage) or urgent intervention indicated | |

| | | Infections and infes | | | |
|---|---|---|---|---|---|
| | | | Grade | - | <u> </u> |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| _aryngitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an inflammatory process in | nvolving the larynx. | • | • | |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder charact | terized by an infectious process invo | lving the lips. | 1 | 1 | |
| Lung infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | terized by an infectious process invo | 1 | I | | 1 |
| Lymph gland infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an infectious process invo | lving the lymph nodes. | <u> </u> | | |
| Mediastinal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an infectious process invo | lving the mediastinum. | | | |
| Meningitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | terized by acute inflammation of the | meninges of the brain and/or spinal | cord. | | |
| Mucosal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an infectious process invo | lving a mucosal surface. | | | |
| Nail infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder charact | terized by an infectious process invo | 1 | Τ | 1 | |
| Otitis externa | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | terized by an infectious process involumptoms include fullness, itching, swe | = | | ive water exposure (swimmer's ea | r infection |
| Otitis media | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an infectious process invo | lving the middle ear. | | | |
| Ovarian infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or antiviral intervention indicated; radiologic or operative | Life-threatening consequences; urgent intervention indicated | Death |

| | 1 | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pancreas infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an infectious process involvi | | | | |
| Papulopustular rash | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | zed by an eruption consisting of pa<br>rash does not present with whiteh | | | | o, and upper |
| Paronychia | Nail fold edema or erythema; disruption of the cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | Surgical intervention or IV antibiotics indicated; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the soft tissues around the nai | l. | <u> </u> | 1 |
| Pelvic infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involvi | ing the pelvic cavity. | 1 | <u> </u> | 1 |
| Penile infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involvi | ing the penis. | T | T | |
| Periorbital infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involvi | | | | |
| Peripheral nerve infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involvi | ing the peripheral nerves. | Т | Т | 1 |
| Peritoneal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involvi | ing the peritoneum. | T | T | |
| Pharyngitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by inflammation of the throat. | 1 | 1 | 1 | 1 |
| Phlebitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | Infections and infestations | | | | |
|---|---|---|---|---|---|
| | | 1 | Grade | I | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | rized by an infectious process in | nvolving the vein. Clinical manifestation | is include erythema, marked disco | omfort, swelling, and induration alo | ng the cour |
| of the infected vein. Pleural infection | | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| ricarar inicotion | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | Death |
| | | antifungal, or antiviral) | radiologic, endoscopic, or | | |
| | | | operative intervention indicated | | |
| Definition: A disorder character | rized by an infectious process in | nvolving the pleura. | T | 1 | |
| Prostate infection | - | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic, endoscopic, or | urgent intervention indicated | |
| | | | operative intervention indicated | | |
| Definition: A disorder characte | rized by an infectious process in | nvolving the prostate gland. | | | |
| Rash pustular | - | Localized; local intervention | IV antibiotic, antifungal, or | - | - |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | | |
| | | antifungal, or antiviral) | radiologic or operative intervention indicated | | |
| Definition: A disorder characte | <br>rized by a circumscribed and ele | l<br>evated skin lesion filled with pus. | Intervention indicated | I | |
| Rhinitis infective | | Localized; local intervention | _ | | |
| Tumino iniconve | | indicated (e.g., topical antibiotic, | | | |
| | | antifungal, or antiviral) | | | |
| Definition: A disorder characte | rized by an infectious process in | nvolving the nasal mucosal. | _ | 1 | |
| Salivary gland infection | - | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., | antiviral intervention indicated; | urgent intervention indicated | |
| | | antibiotic, antifungal, antiviral) | radiologic or operative intervention indicated | | |
| Definition: A disorder characte | rized by an infectious process ir | nvolving the salivary gland. | 1 | I | I |
| Scrotal infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative | | |
| | | | intervention indicated | | |
| | rized by an infectious process in | nvolving the scrotum. | | I | <b>.</b> |
| Sepsis | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: Δ disorder characte | <br>rized by the presence of pathod | enic microorganisms in the blood strea | l<br>om that cause a ranidly progressin | · - | to shock |
| Sinusitis | - Presence of patriog | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Silidollo | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | Death |
| | | antifungal, or antiviral) | radiologic, endoscopic, or | | |
| | | | operative intervention indicated | | |
| | | nvolving the mucous membranes of the | Ĺ | | |
| Skin infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or antiviral intervention indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | indicated | antibiotic, antifuligal, antiviral) | radiologic or operative | argent intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder characte | rized by an infectious process in | nvolving the skin. | | | |
| Small intestine infection | - | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., | antiviral intervention indicated; | urgent intervention indicated | |
| | | antibiotic, antifungal, antiviral) | radiologic or operative intervention indicated | | |
| Definition: A disorder characte | l<br>rized by an infectious process ir | nvolving the small intestine. | 1 | I | I |
| Soft tissue infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative | | |
| | | | intervention indicated | | |
| | rized by an infectious process in | nvolving soft tissues. | <u> </u> | | |
| Splenic infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteria | zed by an infectious process involv | ing the spleen. | Т | 1 | |
| Stoma site infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing a stoma (surgically created op | ening on the surface of the body). | 1 | 1 |
| ooth infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing a tooth. | T | ı | 1 |
| Tracheitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an infectious process involv | ing the trachea. | | | |
| Upper respiratory infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the upper respiratory tract (no | se, paranasal sinuses, pharynx, la | rynx, or trachea). | 1 |
| Urethral infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the urethra. | _ | | |
| Urinary tract infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by an infectious process involv | ing the urinary tract, most commo | nly the bladder and the urethra. | | |
| Uterine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the endometrium. It may exter | . Id to the myometrium and parame | trial tissues. | • |
| Vaginal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an infectious process involv | 1 | | | |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the vulva. | 1 | 1 | |
| Nound infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the wound. | T | | |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ankle fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of damage to affected leg and foot. | o the ankle joint characterized by a | break in the continuity of the ankl | e bone. Symptoms include marke | d discomfort, swelling and difficult | y moving the |
| Aortic injury | - | - | Severe symptoms; limiting self care ADL; disabling; repair or revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | o the aorta. | | | | |
| Arterial injury | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self care ADL; disabling; repair or revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | o an artery. | ' | ' | • | , |
| Biliary anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage or | f bile due to breakdown of a biliary | anastomosis (surgical connection | of two separate anatomic structu | res). | 1 |
| Bladder anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | f urine due to breakdown of a blad | der anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | 1 |
| Bruising | Localized or in a dependent area | Generalized | - | - | - |
| Definition: A finding of injury of the | ne soft tissues or bone characterize | ed by leakage of blood into surrou | nding tissues. | T | I |
| Burn | Minimal symptoms; intervention not indicated | Medical intervention; minimal debridement indicated | Moderate to major debridement or reconstruction indicated | Life-threatening consequences | Death |
| = : | ntegrity to the anatomic site of an adepends on the length and intensi | | | nicals, direct heat, electricity, flame | es and |
| Dermatitis radiation | Faint erythema or dry desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | Death |
| Definition: A finding of cutaneous | s inflammatory reaction occurring a | as a result of exposure to biologica | Illy effective levels of ionizing radia | ation. | |
| Esophageal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an esophagea | l anastomosis (surgical connection | of two separate anatomic structu | res). | |
| Fall | Minor with no resultant injuries; intervention not indicated | Symptomatic; noninvasive intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding of sudden m | ovement downward, usually result | ing in injury. | Γ | Г | 1 |
| Fallopian tube anastomotic leak | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a fallopian tub | e anastomosis (surgical connectio | n of two separate anatomic structu | ures). | |
| Fallopian tube perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated (e.g., organ resection) | Death |
| Definition: A finding of rupture of | the fallopian tube wall. | | 1 | ı | 1 |
| Fracture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic but non-displaced; immobilization indicated | Severe symptoms; displaced or open wound with bone exposure; disabling; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of traumatic | injury to the bone in which the con | tinuity of the bone is broken. | | | |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a gastric anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Gastrointestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a gastrointesti | nal anastomosis (surgical connect | tion of two separate anatomic struc | ctures). | |
| Gastrointestinal stoma necrosis | - | Superficial necrosis; intervention not indicated | Severe symptoms;<br>hospitalization or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of a necrotic | process occurring in the gastroint | estinal tract stoma. | | | |
| Hip fracture | - | Hairline fracture; mild pain;<br>limiting instrumental ADL; non-<br>surgical intervention indicated | Severe pain; hospitalization or intervention indicated for pain control (e.g., traction); operative intervention indicated | Life-threatening consequences; symptoms associated with neurovascular compromise | - |
| Definition: A finding of traumatic | injury to the hip in which the contir | nuity of either the femoral head, fe | moral neck, intertrochanteric or su | btrochanteric regions is broken. | |
| Injury to carotid artery | - | - | Severe symptoms; limiting self<br>care ADL (e.g., transient<br>cerebral ischemia); repair or<br>revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the carotid artery. | | | | |
| Injury to inferior vena cava | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the inferior vena cava. | T | T | T | |
| Injury to jugular vein | - | - | Symptomatic limiting self care ADL; disabling; repair or revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the jugular vein. | T | ı | | |
| Injury to superior vena cava | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; disabling; repair or<br>revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | the superior vena cava. | | | | |
| Intestinal stoma leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | f contents from an intestinal stoma | T T | e surface of the body). | | |
| Intestinal stoma obstruction | - | Self-limited; intervention not indicated | Severe symptoms; IV fluids,<br>tube feeding, or TPN indicated<br>>=24 hrs; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of blockage | of the normal flow of the contents of | of the intestinal stoma. | T | Т | |
| Intestinal stoma site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood leak | age from the intestinal stoma. | | | | |
| Intraoperative arterial injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | an artery during a surgical proce | dure. | | | |
| Intraoperative breast injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | o the breast parenchyma during a | a surgical procedure. | | T | I |
| Intraoperative cardiac injury | - | - | Primary repair of injured organ/structure indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the heart during a surgical proc | edure. | | | |
| Intraoperative ear injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection of injured organ/structure indicated; disabling (e.g., impaired hearing; impaired balance) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the ear during a surgical proced | dure. | | | |
| Intraoperative endocrine injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the endocrine gland during a su | urgical procedure. | | | |
| Intraoperative gastrointestinal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the gastrointestinal system duri | ng a surgical procedure. | | | |
| Intraoperative head and neck injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the head and neck during a sur | gical procedure. | | | |
| Intraoperative hemorrhage | - | - | Postoperative radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of uncontroll | ed bleeding during a surgical pro | cedure. | | | |
| Intraoperative hepatobiliary<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the hepatic parenchyma and/or | biliary tract during a surgical pro | cedure. | | |
| Intraoperative musculoskeletal injury | Primary repair of injured organ/structure indicated of the musculoskeletal system dur | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | | | 0 | l :f- thti | Daath |
| Intraoperative neurological injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | o the nervous system during a su | Ī | | | |
| Intraoperative ocular injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the eye during a surgical proce | dure. | | | |
| Intraoperative renal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the kidney during a surgical pro | ocedure. | | | |
| Intraoperative reproductive tract injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | _ | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of damage to | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the respiratory system during a s | urgical procedure. | | | |
| Intraoperative skin injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the skin during a surgical proced | ure. | | | |
| Intraoperative splenic injury | - | Primary repair of injured organ/structure indicated | Resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | the spleen during a surgical proc | | la " | | <b>5</b> " |
| Intraoperative urinary injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | the urinary system during a surgi | | | | |
| Intraoperative venous injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | a vein during a surgical procedur | re. | | | |
| Kidney anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | f urine due to breakdown of a kidn | ey anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Large intestinal anastomotic eak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the la | rge intestine. | |
| Pancreatic anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a pancreatic a | nastomosis (surgical connection o | f two separate anatomic structures | S). | |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | 1 | | of two separate anatomic structure | • | Dooth |
| Postoperative hemorrhage | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; radiologic, endoscopic, or operative intervention indicated | Transfusion indicated of >=2 units (10 cc/kg for pediatrics) pRBCs beyond protocol specification; urgent radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | occurring after a surgical procedure | | | | _ |
| Postoperative thoracic procedure complication | - | Extubated within 24 - 72 hrs postoperatively | Extubated >72 hrs<br>postoperatively, but before<br>tracheostomy indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A finding of a previous | sly undocumented problem that oc | curs after a thoracic procedure. | 1 | <b>1</b> | 1 |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent after manual<br>reduction; local irritation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental<br>ADL | Severe symptoms; elective operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of protrusion | of the intestinal stoma (surgically | created opening on the surface of | the body) above the abdominal su | urface. | |
| Prolapse of urostomy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Local care or maintenance;<br>minor revision indicated | Dysfunctional stoma; elective operative intervention or major stomal revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of displacement | ent of the urostomy. | 1 | <b>.</b> | 1 | |
| Radiation recall reaction (dermatologic) | Faint erythema or dry desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds | Moist desquamation in areas other than skin folds and creases; bleeding induced by | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous | Death |
| | | and creases; moderate edema | minor trauma or abrasion | bleeding from involved site; skin graft indicated | |
| <del>-</del> | | drugs, especially chemotherapeut ppear after the removal of the pha | <del>-</del> | lowing radiotherapy. The inflamma | tory reaction |
| Rectal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | |
| Definition: A finding of leakage du | ue to breakdown of a rectal anasto | omosis (surgical connection of two | separate anatomic structures). | | |
| Seroma | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; simple aspiration indicated | Symptomatic, elective radiologic or operative intervention indicated | - | - |
| Definition: A finding of tumor-like | collection of serum in the tissues. | ' | ' | ' | ! |
| Small intestinal anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| leak | observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | |
| Definition: A finding of leakage du | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the si | mall bowel. | |
| Spermatic cord anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage du | ue to breakdown of a spermatic co | ord anastomosis (surgical connecti | on of two separate anatomic struc | tures). | Г |
| Spinal fracture | Mild back pain; nonprescription analgesics indicated | Moderate back pain;<br>prescription analgesics<br>indicated; limiting instrumental<br>ADL | Severe back pain;<br>hospitalization or intervention<br>indicated for pain control (e.g.,<br>vertebroplasty); limiting self care<br>ADL; disability | Life-threatening consequences; symptoms associated with neurovascular compromise | Death |
| Definition: A finding of traumatic i | njury to the spine in which the cor | intinuity of a vertebral bone is broke | en. | ! | I |
| Stenosis of gastrointestinal stoma | - | Symptomatic; IV fluids indicated <24 hrs; manual dilation at bedside | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | of the gastrointestinal stoma (surg | gically created opening on the surf | ace of the body). | | |
| Stomal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characterize gastroenterostomy procedure. | ed by a circumscribed, inflammato | ry and necrotic erosive lesion on t | the jejunal mucosal surface close t | to the anastomosis site following a | |
| Tracheal hemorrhage | Minimal bleeding identified on clinical or diagnostic exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding fr | om the trachea. | • | • | • | • |
| Tracheal obstruction | Partial asymptomatic obstruction on examination | Symptomatic (e.g., noisy airway breathing), no respiratory | Stridor; radiologic or endoscopic intervention indicated (e.g., | Life-threatening airway compromise; urgent intervention | Death |
| | (e.g., visual, radiologic or endoscopic) | distress; medical intervention indicated (e.g., steroids); limiting instrumental ADL | stent, laser); limiting self care<br>ADL | indicated (e.g., tracheotomy or intubation) | |
| 56 | of the lumen of the trachea. | • | • | • | i |

| | jury | , poisoning and procedu | | | |
|---|---|---|---|---|---|
| Ad <b>F</b> ( | _ | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Fracheostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood leak | rage from the tracheostomy site. | | _ | | 1 |
| Jreteric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a ureteral ana: | stomosis (surgical connection of two | vo separate anatomic structures). | Т | 1 |
| Jrethral anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a urethral ana | stomosis (surgical connection of two | vo separate anatomic structures). | | |
| Jrostomy leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage o | f contents from a urostomy. | T | T | | |
| Jrostomy obstruction | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; dilation or endoscopic repair or stent placement indicated | Altered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | | | | |
| Urostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding f | rom the urostomy site. | ' | ' | • | , |
| Urostomy stenosis | - | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | of the opening of a urostomy. | | | | |
| Uterine anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a uterine anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Uterine perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a rupture in the uterine wall. | | | | |
| /aginal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a vaginal anas | stomosis (surgical connection of tw | vo separate anatomic structures). | <b>.</b> | 1 |
| /as deferens anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a vas deferens | s anastomosis (surgical connection | n of two separate anatomic structu | res). | |
| Vascular access complication | - | Device dislodgement, blockage,<br>leak, or malposition; device<br>replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including pulmonary embolism or life-threatening thrombus | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Venous injury Definition: A finding of damage t | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self care ADL; repair or revision indicated; disabling | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Wound complication | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound; local care indicated | disruption/dehiscence; primary wound closure or revision by | Hernia with evidence of strangulation; major reconstruction flap, grafting, resection, or amputation indicated | Death |
| Definition: A finding of developm | ent of a new problem at the site of | an existing wound. | T | T | I |
| Wound dehiscence | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of<br>wound with local care;<br>asymptomatic hernia or<br>symptomatic hernia without<br>evidence of strangulation | wound closure or revision by operative intervention indicated | Life-threatening consequences; symptomatic hernia with evidence of strangulation; fascial disruption with evisceration; major reconstruction flap, grafting, resection, or amputation indicated | Death |
| Definition: A finding of separation | of the approximated margins of a | surgical wound. | | | |
| Wrist fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of traumatic | injury to the wrist joint in which the | continuity of a wrist bone is broke | en. | | |
| Injury, poisoning and procedural complications - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Investigations | 3 | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | - | - |
| | · | romboplastin time is found to be g<br>s and disorders, both primary and | reater than the control value. As a related to treatment. | possible indicator of coagulopat | hy, a prolonge |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | ।<br>n increase in the level of alanine a | ı<br>minotransferase (ALT or SGPT) ir | n the blood specimen. | ļ |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of alkaline p | hosphatase in a blood specimen. | ' | 1 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of aspartate | aminotransferase (AST or SGOT | i) in a blood specimen. | ı |
| Blood antidiuretic hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of antidiuretic horm | one in the blood specimen. | 1 | |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormally high level of bilirubin | in the blood. Excess bilirubin is as | ssociated with jaundice. | |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of corticotrop | nin in a blood specimen. | | |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | ,<br>bnormal levels of gonadotrophin h | ormone in a blood specimen. | ' | 1 |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of prolactin hormor | ne in a blood specimen. | ' | ' |
| Carbon monoxide diffusing capacity decreased | up, a decrease of 3 - 5 units<br>(ml/min/mm Hg) below the<br>baseline value | 6 - 8 units below LLN; for follow-<br>up, an asymptomatic decrease<br>of >5 - 8 units (ml/min/mm Hg)<br>below the baseline value | Asymptomatic decrease of >8 units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., >Grade 2 hypoxia or >Grade 2 or higher dyspnea) | - | - |
| | | a decrease in the lung capacity | | | |
| Cardiac troponin I increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | | Levels consistent with myocardial infarction as defined by the manufacturer | | |
| Definition: A laboratory test result | | of cardiac troponin I in a biologica | I specimen. | I | |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| Definition: A laboratory test result | · · | ।<br>of cardiac troponin T in a biologica | al specimen. | • | • |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 10e9="" 500="" <lln="" l<="" mm3;="" td="" x=""><td>&lt;500 - 200/mm3; &lt;0.5 - 0.2 x<br/>10e9 /L</td><td>&lt;200 - 50/mm3; &lt;0.2 x 0.05 -<br/>10e9 /L</td><td>&lt;50/mm3; &lt;0.05 x 10e9 /L</td><td>-</td></lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of CD4 lymph | ocytes in a blood specimen. | | |
| Cholesterol high | >ULN - 300 mg/dL; >ULN - 7.75<br>mmol/L | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | >400 - 500 mg/dL; >10.34 -<br>12.92 mmol/L | >500 mg/dL; >12.92 mmol/L | - |
| Definition: A finding based on lab | oratory test results that indicate hi | gher than normal levels of choles | erol in a blood specimen. | | |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN n increase in levels of creatine pho | >5 x ULN - 10 x ULN | >10 x ULN | - |

| | | Investigations | 3 | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Creatinine increased | >1 - 1.5 x baseline; >ULN - 1.5 x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of creatinine in a b | iological specimen. | | |
| Ejection fraction decreased | - used when the amount of blood sig | - 40%; 10 - 19% drop from baseline | Resting ejection fraction (EF) 39 - 20%; >20% drop from baseline ion of the heart is compared to the | <20% | - |
| contraction. | uted when the amount of blood eje | ected during a ventricular contracti | ion of the heart is compared to the | amount that was present prior to | uie |
| Electrocardiogram QT corrected interval prolonged | | QTc 481 - 500 ms | 1 | QTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | - |
| - | dysrhythmia characterized by an a | | | | |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50%<br>decrease from baseline | <0.5 - 0.25 x LLN or 50 - <75% decrease from baseline | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of fibrinogen i | n a blood specimen. | | |
| Forced expiratory volume decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| Definition: A finding based on tes | t results that indicate a relative de | crease in the fraction of the forced | vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate hi | gher than normal levels of the enz | zyme gamma-glutamyltransferase | in the blood specimen. GGT (gam | ıma- |
| glutamyltransferase ) catalyzes ti | ne transfer of a gamma glutamyl g | roup from a gamma glutamyl pept | ide to another peptide, amino acid | s or water. | |
| Growth hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | onormal levels of growth hormone | in a biological specimen. | ı | 1 |
| Haptoglobin decreased | <lln< td=""><td>-</td><td>-</td><td>-</td><td>-</td></lln<> | - | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of haptoglobir | in a blood specimen. | I | ı |
| Hemoglobin increased | Increase in >0 - 2 gm/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | - | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of hemoglobin in a | 1 | | |
| INR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5<br>times above baseline if on<br>anticoagulation | >2.5 x ULN; >2.5 times above baseline if on anticoagulation | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the ratio of the patier | nt's prothrombin time to a control s | ample in the blood. | T |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of lipase in | a biological specimen. | T | T |
| Lymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <800 - 500/mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of lymphocyte | es in a blood specimen. | <b>I</b> | 1 |
| Lymphocyte count increased | - | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormal increase in the numbe | r of lymphocytes in the blood, effu | sions or bone marrow. | 1 |
| Neutrophil count decreased | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of neutrophils | s in a blood specimen. | <b>I</b> | |
| Pancreatic enzymes decreased | <lln and="" asymptomatic<="" td=""><td>Increase in stool frequency, bulk, or odor; steatorrhea</td><td>Sequelae of absorption deficiency</td><td>-</td><td>-</td></lln> | Increase in stool frequency, bulk, or odor; steatorrhea | Sequelae of absorption deficiency | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of pancreatic | enzymes in a biological specimen | | |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" -<br="" 75,000="" <lln="" mm3;="">75.0 x 10e9 /L</lln> | <75,000 - 50,000/mm3; <75.0 - 50.0 x 10e9 /L | <50,000 - 25,000/mm3; <50.0 - 25.0 x 10e9 /L | <25,000/mm3; <25.0 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate ar | n increase in the levels of amylase | in a serum specimen. | | |
| Urine output decreased | - | - | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | - |
| Definition: A finding based on tes | t results that indicate urine produc | tion is less relative to previous ou | tput. | | |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value;<br>limiting instrumental ADL | <50% of predicted value;<br>limiting self care ADL | - | - |
| Definition: A finding based on pul value. | lmonary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | uum inhalation) when compared to | the predicted |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characterized | d by an increase in overall body we | ·<br>eight; for pediatrics, greater than t | he baseline growth curve. | • | ' |
| Weight loss | 5 to <10% from baseline;<br>intervention not indicated | 10 - <20% from baseline;<br>nutritional support indicated | >=20% from baseline; tube feeding or TPN indicated | - | - |
| Definition: A finding characterized | d by a decrease in overall body we | eight; for pediatrics, less than the b | paseline growth curve. | | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <3000 - 2000/mm3; <3.0 - 2.0 x<br>10e9 /L | <2000 - 1000/mm3; <2.0 - 1.0 x<br>10e9 /L | <1000/mm3; <1.0 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate ar | n decrease in number of white blo | od cells in a blood specimen. | | |
| Investigations - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Metabolism and nutrition | | | |
|---|---|---|---|---|---|
| | | _ | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | Death |
| Definition: A disorder characterize | ed by abnormally high acidity (high | n hydrogen-ion concentration) of the | he blood and other body tissues. | | |
| Alcohol intolerance | <del>-</del><br> - | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize comiting, indigestion and headact | - | the adverse effects of alcohol, whi | ich can include nasal congestion, s | skin flushes, heart dysrhythmias, r | nausea, |
| Alkalosis | pH >normal, but <=7.5 | - | pH >7.5 | Life-threatening consequences | Death |
| Definition: A disorder characterize | ed by abnormally high alkalinity (lo | ow hydrogen-ion concentration) of | the blood and other body tissues. | | |
| Anorexia | Loss of appetite without alteration in eating habits | Oral intake altered without significant weight loss or malnutrition; oral nutritional supplements indicated | Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); tube feeding or TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a loss of appetite. | Г | T | Т | |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated <24 hrs | IV fluids or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| ا<br>Definition: A disorder characterize | _ | l<br>h the hody. It is usually caused by | severe diarrhea, vomiting or diaph | l<br>noresis | l |
| Glucose intolerance | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an inability to properly metal | bolize glucose. | | | |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of<br>>11.5 - 12.5 mg/dL; >2.9 - 3.1<br>mmol/L; lonized calcium >1.5 -<br>1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; lonized calcium >1.8 mmol/L; life-threatening consequences | Death |
| ا<br>Definition: A disorder characterize | ed by laboratory test results that ir | dicate an elevation in the concen | tration of calcium (corrected for alk | oumin) in blood. | 1 |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8.9 mmol/L | Fasting glucose value >160 -<br>250 mg/dL; Fasting glucose<br>value >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characterize ntolerance. | ed by laboratory test results that in | ndicate an elevation in the concen | tration of blood sugar. It is usually | an indication of diabetes mellitus | or glucose |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize<br>the use of diuretic drugs. | ed by laboratory test results that ir | ndicate an elevation in the concen | tration of potassium in the blood; a | associated with kidney failure or so | metimes |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23 mmol/L | - | >3.0 - 8.0 mg/dL; >1.23 - 3.30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | ed by laboratory test results that ir | ndicate an elevation in the concen | tration of magnesium in the blood | | |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | ed by laboratory test results that in | ndicate an elevation in the concen | tration of sodium in the blood. | | |
| Hypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42 mmol/L | >300 mg/dL - 500 mg/dL; >3.42<br>mmol/L - 5.7 mmol/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4 mmol/L | >1000 mg/dL; >11.4 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | ed by laboratory test results that ir | ndicate an elevation in the concen | tration of triglyceride concentration | in the blood. | |
| Hyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic<br>consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences | >10 mg/dL; >0.59 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characterize | ed by laboratory test results that in | ndicate an elevation in the concen | tration of uric acid. | | |
| Hypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypocalcemia | Corrected serum calcium of<br><lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln -<br="">1.0 mmol/L</lln></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 - 6.0 mg/dL; <1.75 - 1.5<br>mmol/L; lonized calcium <0.9 -<br>0.8 mmol/L; hospitalization<br>indicated | Corrected serum calcium of<br><6.0 mg/dL; <1.5 mmol/L;<br>lonized calcium <0.8 mmol/L;<br>life-threatening consequences | Death |
| Definition: A disorder character | rized by laboratory test results that in | ndicate a low concentration of calc | ium (corrected for albumin) in the | blood. | |
| Hypoglycemia | <lln -="" 3.0="" 55="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;55 - 40 mg/dL; &lt;3.0 - 2.2<br/>mmol/L</td><td>&lt;40 - 30 mg/dL; &lt;2.2 - 1.7<br/>mmol/L</td><td>&lt;30 mg/dL; &lt;1.7 mmol/L; life-<br/>threatening consequences;<br/>seizures</td><td>Death</td></lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7<br>mmol/L | <30 mg/dL; <1.7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| Definition: A disorder character | rized by laboratory test results that in | ndicate a low concentration of gluc | ose in the blood. | | |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><pre><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" pre="" symptomatic;=""></lln></pre></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <pre><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" pre="" symptomatic;=""></lln></pre> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening consequences | Death |
| Definition: A disorder character | rized by laboratory test results that ir | ndicate a low concentration of pota | assium in the blood. | | |
| Hypomagnesemia | <lln -="" 0.5<br="" 1.2="" <lln="" dl;="" mg="">mmol/L</lln> | <1.2 - 0.9 mg/dL; <0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3 mmol/L | <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences | Death |
| Definition: A disorder character | rized by laboratory test results that ir | ndicate a low concentration of mag | nesium in the blood. | _ | |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder character | rized by laboratory test results that ir | ndicate a low concentration of sodi | ium in the blood. | | |
| Hypophosphatemia | <lln -="" 0.8<br="" 2.5="" <lln="" dl;="" mg="">mmol/L</lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6 mmol/L | <2.0 - 1.0 mg/dL; <0.6 - 0.3 mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder character | rized by laboratory test results that ir | ndicate a low concentration of pho | sphates in the blood. | | |
| Iron overload | - | Moderate symptoms; intervention not indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by accumulation of iron in the t | issues. | | | |
| Obesity | - | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | - |
| Definition: A disorder character | rized by having a high amount of boo | dy fat. | | | |
| Tumor lysis syndrome | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by metabolic abnormalities that | result from a spontaneous or the | rapy-related cytolysis of tumor cell | S. | |
| Metabolism and nutrition disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | - | 2 | Grade 3 | 4 | 5 |
|---|---|---|---|---|---|
| Abdominal soft tissue necrosis | - | | • | 7 | |
| Definition: A disorder characteriz | | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a necrotic process occurring | in the soft tissues of the abdomir | nal wall. | | |
| Arthralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in a joint. | T | T | |
| Arthritis | Mild pain with inflammation, erythema, or joint swelling | Moderate pain associated with signs of inflammation, erythema, or joint swelling; limiting instrumental ADL | Severe pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inflammation involving a joir | ıt. | | | |
| Avascular necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by necrotic changes in the bond the destruction of the bone struc | • | od supply. Most often affecting the | epiphysis of the long bones, the n | ecrotic |
| Back pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the back region. | _ | _ | |
| Bone pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the bones. | 1 | 1 | |
| Buttock pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | ed by marked discomfort sensation | | | | |
| Chest wall pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | ed by marked discomfort sensation | n in the chest wall region. | | | |
| Exostosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by non-neoplastic overgrowth c | of bone. | • | • | |
| Fibrosis deep connective tissue | Mild induration, able to move skin parallel to plane (sliding) and perpendicular to skin (pinching up) | Moderate induration, able to slide skin, unable to pinch skin; limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| | ed by fibrotic degeneration of the o | · · | | | |
| Flank pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n on the lateral side of the body in | the region below the ribs and about | ove the hip. | |
| Generalized muscle weakness | Symptomatic; weakness perceived by patient but not evident on physical exam | Symptomatic; weakness evident<br>on physical exam; weakness<br>limiting instrumental ADL | Weakness limiting self care<br>ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f muscles in multiple anatomic sit | es. | | |
| Growth suppression | Reduction in growth velocity by<br>10 - 29% ideally measured over<br>the period of a year | Reduction in growth velocity by 30 - 49% ideally measured over the period of a year or 0 - 49% reduction in growth from the baseline growth curve | Reduction in growth velocity of >=50% ideally measured over the period of a year | - | - |

| Figure Part | | | loskeletal and connectiv | Grade | | |
|---|---|---|---|---|---|---|
| Local wound carer, medical infervention indicated (e.g., a disorder characterized by a necrotic process occurring in the soft fasues of the flusten of dispersable cobservations out of dispersable cobservations of dispersable cobservations out of dispersable cobser | Adverse Event | 1 | 2 | | 4 | 5 |
| Joint ange of motion decreased recording to the extension of the disposate characterized by a cerease in place of the provided | | - | Local wound care; medical intervention indicated (e.g., dressings or topical | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap | Life-threatening consequences; | |
| diagnosis observations only; intervention not indicated by accessive fluid in a joint, usually as a result of joint inflammation. Joint range of motion decreased Service (1964) (and point) of the properties of | Definition: A disorder characterize | ed by a necrotic process occurring | in the soft tissues of the head. | | | |
| motion/, decreased ROM limiting antitletic activity Definition: A disorder characterized by a decrease in joint flooibility of any joint. Rotation < | Joint effusion | diagnostic observations only; | | care ADL; elective operative | - | - |
| Initiality and all series care ADL; disabling instrumental ADL initiality and series care ADL; disabling initiality and series and series activity of any joint. Rotation <a 2"="" href="#package=">Rotation or decreases of the series of the seri</a> | | | | | | |
| Rotation - 680 degrees to right or new flexion between 60 - 70 degrees left; 60 degrees of flexion left; 60 degrees of the flexion left; 60 degrees of | Joint range of motion decreased | motion); decreased ROM | · | | - | - |
| Definition: A disorder characterized by a decrease in flexibility of a cervical spine of the floor to pick up a very light object from the floor floor to pick up a very light object or death of the very light object floor to pick up a very light object or death of the very light object or death of the very light object floor to pick up a very light object or death of the very light object or death of the very limb floor of the very limb floor floo | Definition: A disorder characterize | ed by a decrease in joint flexibility | of any joint. | | | |
| Joint range of motion decreased lumbar spine (ROM) in lumbar spine activity bending to the floor to pick up a very light object but able to do athletic activity and spine; required to pick up a very light object from the floor of pick up a very light object from the floor of pick up a very light object from the floor of pick up a very light object from the floor of pick up a very light object from the floor of diagnostic observations only; intervention on indicated of diagnostic observations only; intervention on indicated or diagnostic observations only; intervention on or the spine. Definition: A disorder characterized by a reduction in the strength of the unsueles on the left side of the body. Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the ower limb unsueles. Symptomatic; perceived by symptomatic; perceived by symptomatic; evident on physical | Joint range of motion decreased cervical spine | | | segments with no C-spine | - | - |
| tumbar spine the floor to pick up a very light object but able to do athletic activity should be to do athletic activity should be to do athletic activity should be to do athletic activity should be to do athletic activity should be to be to be seen to floor to pick up a very light object from the floor should be segments with not L-spine flexion (e.g., unable to reach to floor to pick up a very light object) should be segments with not L-spine flexion (e.g., unable to reach to floor to pick up a very light object) should be segments with not L-spine flexion (e.g., unable to reach to floor to pick up a very light object) should be segments with not L-spine flexion (e.g., unable to reach to floor to pick up a very light object) should be segments with not L-spine flexion (e.g., unable to reach to floor to pick up a very light object from the floor should be segments with not L-spine flexion (e.g., unable to reach to floor to pick up a very light object) should be segments with not L-spine flexion (e.g., unable to reach to floor to pick up a very light object from the floor should be segments with not L-spine flexion (e.g., unable to reach to flexion to pick up a very light object from the floor should be segments with not L-spine flexion (e.g., unable to reach to flexion flexion flexio | Definition: A disorder characterize | ed by a decrease in flexibility of a | cervical spine joint. | T | T | |
| Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by an abnormal increase in the curvature of the thoracic portion of the spine. Lordosis Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by an abnormal increase in the curvature of the thoracic portion of the spine. Lordosis Asymptomatic; clinical or diagnostic observations only; intervention not indicated Instrumental ADL Severe accentuation; limiting self care ADL Severe accentuation; operative intervention indicated; limiting instrumental ADL Severe accentuation; operative intervention indicated; limiting self care ADL Severe accentuation; operative intervention indicated; limiting self care ADL Severe accentuation; operative intervention indicated; limiting self care ADL Severe accentuation; operative intervention indicated; limiting self care ADL Severe accentuation; operative intervention indicated; limiting self care ADL Limiting self care ADL; disabling ophysical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Muscle weakness trunk Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Symptomatic; perceived by pati | = | the floor to pick up a very light object but able to do athletic | (ROM) in lumbar spine; requires a reaching aid to pick up a very | associated with symptoms of<br>ankylosis or fused over multiple<br>segments with no L-spine<br>flexion (e.g., unable to reach to<br>floor to pick up a very light | - | - |
| diagnostic observations only; instrumental ADL instrumental ADL self-care ADL self-car | Definition: A disorder characterize | ed by a decrease in flexibility of a | lumbar spine joint. | | | |
| Asymptomatic; clinical or diagnostic observations only; intervention not indicated; limiting instrumental ADL Definition: A disorder characterized by an abnormal increase in the curvature of the lumbar portion of the spine. Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the left side of the body. Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb muscles. Muscle weakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb muscles. Muscle weakness trunk Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Symptomatic; evident on physical exam; limiting instrumental ADL Limiting self care ADL; disabling physical exam; limiting instrumental ADL Limiting self care ADL; disabling | Kyphosis | diagnostic observations only; | | intervention indicated; limiting | - | - |
| diagnostic observations only; instrumental ADL intervention indicated; limiting self care ADL Definition: A disorder characterized by an abnormal increase in the curvature of the lumbar portion of the spine. Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb whise lewakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb whise lewakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb muscles. Muscle weakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on physical exam; limiting instrumental ADL Limiting self care ADL; disabling | Definition: A disorder characterize | ed by an abnormal increase in the | curvature of the thoracic portion of | of the spine. | <b>.</b> | |
| Muscle weakness left-sided | Lordosis | diagnostic observations only; | _ | intervention indicated; limiting | - | - |
| patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the left side of the body. Muscle weakness lower limb Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb muscles. Muscle weakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Muscle weakness trunk Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on Limiting self care ADL; disabling | Definition: A disorder characterize | ed by an abnormal increase in the | curvature of the lumbar portion of | f the spine. | | |
| Muscle weakness lower limb Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb muscles. Muscle weakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Muscle weakness trunk Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Symptomatic; evident on Limiting self care ADL; disabling | Muscle weakness left-sided | patient but not evident on | physical exam; limiting | Limiting self care ADL; disabling | - | - |
| patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the lower limb muscles. Muscle weakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Muscle weakness trunk Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on Limiting self care ADL; disabling | Definition: A disorder characterize | ed by a reduction in the strength o | f the muscles on the left side of th | e body. | T | |
| Muscle weakness right-sided Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; evident on physical exam; limiting instrumental ADL Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on physical exam; limiting instrumental ADL Limiting self care ADL; disabling | Muscle weakness lower limb | patient but not evident on | physical exam; limiting | Limiting self care ADL; disabling | - | - |
| patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles on the right side of the body. Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on Physical exam; limiting self care ADL; disabling Physical exam; limiting self care ADL; disabling Physical exam; limiting Physical ex | Definition: A disorder characterize | ed by a reduction in the strength o | f the lower limb muscles. | T | T | |
| Muscle weakness trunk Symptomatic; perceived by patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; evident on physical exam; limiting instrumental ADL Limiting self care ADL; disabling | Muscle weakness right-sided | patient but not evident on | physical exam; limiting | Limiting self care ADL; disabling | - | - |
| patient but not evident on physical exam; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the trunk muscles. Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on Limiting self care ADL; disabling | Definition: A disorder characterize | ed by a reduction in the strength o | f the muscles on the right side of t | the body. | | |
| Muscle weakness upper limb Symptomatic; perceived by Symptomatic; evident on Limiting self care ADL; disabling | Muscle weakness trunk | patient but not evident on | physical exam; limiting | Limiting self care ADL; disabling | - | - |
| | Definition: A disorder characterize | ed by a reduction in the strength o | f the trunk muscles. | T | | |
| physical exam instrumental ADL | Muscle weakness upper limb | patient but not evident on | physical exam; limiting | Limiting self care ADL; disabling | - | - |

| | Muscu | loskeletal and connectiv | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Musculoskeletal deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis (e.g.,<br>shoe insert) or covered by<br>clothing | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>clothing; disabling | - | - |
| Definition: A disorder characteriz | ed by of a malformation of the mus | sculoskeletal system. | | | |
| Myalgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n originating from a muscle or gro | up of muscles. | | |
| Myositis | Mild pain | Moderate pain associated with weakness; pain limiting instrumental ADL | Pain associated with severe weakness; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inflammation involving the s | keletal muscles. | | | |
| Neck pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the neck area. | T | | |
| Neck soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the neck. | T | | |
| Osteonecrosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the bone of the mandible. | | | |
| Osteoporosis | Radiologic evidence of<br>osteoporosis or Bone Mineral<br>Density (BMD) t-score -1 to -2.5<br>(osteopenia); no loss of height<br>or intervention indicated | BMD t-score <-2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >=2 cm;<br>hospitalization indicated; limiting<br>self care ADL | - | - |
| Definition: A disorder characteriz composition), resulting in increas | ed by reduced bone mass, with a | decrease in cortical thickness and | in the number and size of the trab | eculae of cancellous bone (but no | rmal chemic |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the upper or lower extremities | i. | | |
| Pelvic soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a necrotic process occurring | in the soft tissues of the pelvis. | T | | |
| Scoliosis | <20 degrees; clinically undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward flexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a malformed, lateral curvatu | re of the spine. | T | | |
| Soft tissue necrosis lower limb | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a necrotic process occurring | in the soft tissues of the lower ex | tremity. | | |
| Soft tissue necrosis upper limb | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| | | | ktremity. | | |
| | Muscu | loskeletal and connectiv | e tissue disorders | | | | | |
|---|---|---|---|---|---|--|--|--|
| | Grade | | | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 | | | |
| Superficial soft tissue fibrosis | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to slide skin, unable to pinch skin; limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death | | | |
| Definition: A disorder characteriz | ed by fibrotic degeneration of the | superficial soft tissues. | | | | | | |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring small bites, soft foods or purees | Decreased ROM with inability to adequately aliment or hydrate orally | - | - | | | |
| Definition: A disorder characteriz | ed by lack of ability to open the mo | outh fully due to a decrease in the | range of motion of the muscles of | mastication. | | | | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 - 5 cm; shoe lift indicated; limiting instrumental ADL | Severe length discrepancy >5 cm; limiting self care ADL; disabling; operative intervention indicated | - | - | | | |
| Definition: A disorder characteriz | ed by of a discrepancy between th | e lengths of the lower or upper ex | tremities. | | | | | |
| Musculoskeletal and connective tissue disorder - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death | | | |

| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Leukemia secondary to | - | - | - | Present | Death |
| oncology chemotherapy | | | | | |
| Definition: A disorder characteriz | ed by leukemia arising as a result | of the mutagenic effect of chemo | therapy agents. | | |
| Myelodysplastic syndrome | - | - | - | Life-threatening consequences; | Death |
| | | | | urgent intervention indicated | |
| Definition: A disorder characteriz | ed by insufficiently healthy hemata | poietic cell production by the bor | e marrow. | • | |
| Treatment related secondary | - | - | Non life-threatening secondary | Acute life-threatening secondary | Death |
| malignancy | | | malignancy | malignancy; blast crisis in | |
| | | | | leukemia | |
| Definition: A disorder characteriz | ed by development of a malignand | cy most probably as a result of tre | atment for a previously existing ma | alignancy. | |
| Tumor pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder characteriz | ed by marked discomfort from a ne | eoplasm that may be pressing on | a nerve, blocking blood vessels, ir | flamed or fractured from metastas | is. |
| Neoplasms benign, malignant | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| and unspecified (incl cysts and | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| polyps) - Other, specify | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| Nervous system disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abducens nerve disorder | Asymptomatic; clinical or diagnostic observations only; | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| | intervention not indicated | | | | |
| Definition: A disorder characteri | zed by involvement of the abducen | s nerve (sixth cranial nerve). | | | |
| Accessory nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | | | | |
| | zed by involvement of the accessor | İ | <u> </u> | | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by involvement of the acoustic | nerve (eighth cranial nerve). | ' | ' | |
| Akathisia | Mild restlessness or increased | Moderate restlessness or | Severe restlessness or | - | - |
| | motor activity | increased motor activity; limiting instrumental ADL | increased motor activity; limiting self care ADL | | |
| Definition: A disorder characteri | zed by an uncomfortable feeling of | inner restlessness and inability to | stay still; this is a side effect of so | me psychotropic drugs. | 1 |
| Amnesia | Mild; transient memory loss | Moderate; short term memory loss; limiting instrumental ADL | Severe; long term memory loss; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by systematic and extensive lo | ss of memory. | | | |
| Aphonia | - | - | Voicelessness; unable to speak | - | - |
| Definition: A disorder characteri | zed by the inability to speak. It may | result from injuries to the vocal co | ords or may be functional (psychog | genic). | |
| Arachnoiditis | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by inflammation of the arachno | id membrane and adjacent subara | achnoid space. | T | |
| Ataxia | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; intervention not indicated | instrumental ADL | care ADL; mechanical assistance indicated | | |
| Definition: A disorder characteri | zed by lack of coordination of musc | le movements resulting in the imp | 1 | Intary activities | l |
| Brachial plexopathy | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | | I |
| Statistical precopatity | diagnostic observations only;<br>intervention not indicated | instrumental ADL | care ADL | | |
| Definition: A disorder characteri | zed by regional paresthesia of the b | orachial plexus, marked discomfor | t and muscle weakness, and limite | ed movement in the arm or hand. | , |
| Central nervous system | Asymptomatic; clinical or | Moderate symptoms; | Severe symptoms; medical | Life-threatening consequences; | Death |
| necrosis | diagnostic observations only; intervention not indicated | corticosteroids indicated | intervention indicated | urgent intervention indicated | |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the brain and/or spinal cord | I | I | 1 |
| Cerebrospinal fluid leakage | Post-craniotomy: asymptomatic; | Post-craniotomy: moderate | Severe symptoms; medical | Life-threatening consequences; | Death |
| | Post-lumbar puncture: transient | symptoms; medical intervention | intervention indicated | urgent intervention indicated | _ 5001 |
| | headache; postural care | indicated; Post-lumbar | | | |
| | indicated | puncture: persistent moderate symptoms; blood patch | | | |
| Definition: A disorder characteri | <br>zed by loss of cerebrospinal fluid in | indicated | I | I | I |
| Cognitive disturbance | Mild cognitive disability; not | Moderate cognitive disability; | Severe cognitive disability; | | |
| ooganiivo aistarbario <del>c</del> | interfering with work/school/life | interfering with work/school/life | significant impairment of | | |
| | performance; specialized | performance but capable of | work/school/life performance | | |
| | educational services/devices | independent living; specialized | | | |
| | not indicated | resources on part time basis indicated | | | |
| Definition: A disorder characteri | l<br>zed by a conspicuous change in co | 1 | I | I | Į. |
| Concentration impairment | Mild inattention or decreased | Moderate impairment in | Severe impairment in attention | _ | l _ |
| osoonaaaon impailment | level of concentration | attention or decreased level of | or decreased level of | | |
| | | concentration; limiting | concentration; limiting self care | | |
| | 1 | instrumental ADL | ADL | i | 1 |

| Nervous system disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to stimuli; limiting instrumental ADL | Difficult to arouse | Life-threatening consequences | Death |
| Definition: A disorder characte | rized by a decrease in ability to perc | eive and respond. | _ | | |
| Dizziness | Mild unsteadiness or sensation of movement | Moderate unsteadiness or sensation of movement; limiting instrumental ADL | Severe unsteadiness or sensation of movement; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a disturbing sensation of lig | htheadedness, unsteadiness, gidd | iness, spinning or rocking. | | |
| Dysarthria | Mild slurred speech | Moderate impairment of articulation or slurred speech | Severe impairment of articulation or slurred speech | - | - |
| Definition: A disorder characte | rized by slow and slurred speech res | sulting from an inability to coordina | te the muscles used in speech. | Т | |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| Definition: A disorder characte | rized by distortion of sensory percep | tion, resulting in an abnormal and | unpleasant sensation. | 1 | |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in diet (e.g., oral supplements); noxious or unpleasant taste; loss of taste | - | - | - |
| Definition: A disorder characte | rized by abnormal sensual experience | ce with the taste of foodstuffs; it ca | n be related to a decrease in the | sense of smell. | |
| Dysphasia | Awareness of receptive or expressive characteristics; not impairing ability to communicate | Moderate receptive or expressive characteristics; impairing ability to communicate spontaneously | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly | - | - |
| Definition: A disorder characte | rized by impairment of verbal comm | unication skills, often resulting from | n brain damage. | ı | 1 |
| Edema cerebral | - | - | - | Life-threatening consequences; urgent intervention indicated | - |
| Definition: A disorder characte | rized by swelling due to an excessive | e accumulation of fluid in the brain | | | |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a pathologic process involvi | ng the brain. | I | T | |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary movements; limiting instrumental ADL | Severe involuntary movements or torticollis; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by abnormal, repetitive, involur | ntary muscle movements, frenzied | speech and extreme restlessness | i. | |
| Facial muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a reduction in the strength of | of the facial muscles. | | | |
| Facial nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by involvement of the facial ne | rve (seventh cranial nerve). | | | |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by involvement of the glossoph | naryngeal nerve (ninth cranial nerv | e). | | |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in various parts of the head | not confined to the area of distrib | ution of any nerve. | |
| Hydrocephalus | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; intervention not indicated | Severe symptoms or neurological deficit; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal increase of ce | rebrospinal fluid in the ventricles o | f the brain. | | 1 |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for sleep | Severe increased need for sleep | - | - |
| Definition: A disorder abarests | rized by characterized by excessive | sleepiness during the daytime. | | • | • |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| lypoglossal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| efinition: A disorder characterize | zed by involvement of the hypoglos | sal nerve (twelfth cranial nerve). | _ | | |
| ntracranial hemorrhage | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteriz | zed by bleeding from the cranium. | I | Ι | T | |
| schemia cerebrovascular | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | - | - | - |
| efinition: A disorder characteriz amage. | zed by a decrease or absence of bl | ood supply to the brain caused by | obstruction (thrombosis or embol | ism) of an artery resulting in neuro | logical |
| Vth nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| efinition: A disorder characteriz | zed by involvement of the trochlear | nerve (fourth cranial nerve). | Т | T | |
| ethargy | Mild symptoms; reduced alertness and awareness | Moderate symptoms; limiting instrumental ADL | - | - | - |
| efinition: A disorder characteriz | zed by a decrease in consciousnes | s characterized by mental and phy | ysical inertness. | T | 1 |
| _eukoencephalopathy | Asymptomatic; small focal T2/FLAIR hyperintensities; involving periventricular white matter or <1/3 of susceptible areas of cerebrum +/- mild increase in subarachnoid space (SAS) and/or mild ventriculomegaly | Moderate symptoms; focal T2/FLAIR hyperintensities, involving periventricular white matter extending into centrum semiovale or involving 1/3 to 2/3 of susceptible areas of cerebrum +/- moderate increase in SAS and/or moderate ventriculomegaly | Severe symptoms; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving 2/3 or more of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Life-threatening consequences; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Death |
| Definition: A disorder characteriz | zed by diffuse reactive astrocytosis | with multiple areas of necrotic for | i<br>i without inflammation. | | ı |
| Memory impairment | Mild memory impairment | Moderate memory impairment;<br>limiting instrumental ADL | Severe memory impairment;<br>limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by a deterioration in memory fu | inction. | | | |
| /leningismus | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterization | zed by neck stiffness, headache, ar | nd photophobia resulting from irrita | ation of the cerebral meninges. | 1 | 1 |
| Novements involuntary | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| | zed by uncontrolled and purposeles | ss movements. | Ι | T | 1 |
| <i>Myelitis</i> | Asymptomatic; mild signs (e.g.,<br>Babinski's reflex or Lhermitte's<br>sign) | Moderate weakness or sensory loss; limiting instrumental ADL | Severe weakness or sensory loss; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteriz | zed by inflammation involving the s | , | 1 | marked discomfort and incontiner | nce. |
| leuralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| efinition: A disorder characteriz | zed by intense painful sensation ald | I - | <u> </u> | T | |
| ystagmus | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| efinition: A disorder characteriz | red by involuntary movements of the | ne eyeballs. | I | T | |
| Oculomotor nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the oculomo | tor nerve (third cranial nerve). | | | |
| Olfactory nerve disorder | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Sofinition: A disorder abaracteri- | zed by involvement of the olfactory | nerve (first cranial nerve). | | | |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz are experienced in the absence of | | ensory neurons resulting in abnorr | mal cutaneous sensations of tinglir | ng, numbness, pressure, cold, and | warmth that |
| Peripheral motor neuropathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; assistive device indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz Peripheral sensory neuropathy | Asymptomatic; loss of deep tendon reflexes or paresthesia | n of the peripheral motor nerves. Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation or degeneratio | n of the peripheral sensory nerves | S. | T | |
| Phantom pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort related to | a limb or an organ that is remove | ed from or is not physically part of | the body. | |
| Presyncope | - | Present (e.g., near fainting) | - | - | - |
| Definition: A disorder characteriz | ed by an episode of lightheadedne | ess and dizziness which may prec | ede an episode of syncope. | | |
| Pyramidal tract syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by dysfunction of the corticospi<br>and a decrease in fine motor coord | | l cord. Symptoms include an incre | ease in the muscle tone in the lowe | er extremities, |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting instrumental ADL; medical intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz connecting nerve root. | ed by inflammation involving a ner | ve root. Patients experience mark | ed discomfort radiating along a ne | erve path because of spinal pressu | re on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by paralysis of the recurrent lar | yngeal nerve. | | | |
| Reversible posterior leukoencephalopathy syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; abnormal imaging studies; limiting instrumental ADL | Severe symptoms; very<br>abnormal imaging studies;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | | = | | indings of posterior leukoencephal<br>s an acute or subacute reversible o | - |
| Seizure | Brief partial seizure; no loss of consciousness | Brief generalized seizure | Multiple seizures despite medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characteriz | ed by a sudden, involuntary skelet | al muscular contractions of cerebi | ral or brain stem origin. | T | |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort in the fac | ce, between the eyes, or upper tee | eth originating from the sinuses. | | |
| Somnolence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stupor | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by characterized by excessive | sleepiness and drowsiness. | Ī | | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle tone and increase in resistance through range of motion | Severe increase in muscle tone and increase in resistance through range of motion | Life-threatening; unable to move active or passive range of motion | Death |
| Definition: A disorder characteriz disturbances. | ed by increased involuntary muscl | e tone that affects the regions inte | erfering with voluntary movement. | It results in gait, movement, and sp | peech |
| Stroke | Asymptomatic or mild neurologic deficit; radiographic findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a sudden loss of sensory fu | nction due to an intracranial vascu | ılar event. | | |
| Syncope | - | - | Fainting; orthostatic collapse | - | - |
| Definition: A disorder characteriz | ed by spontaneous loss of conscio | ousness caused by insufficient blo | od supply to the brain. | | |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Transient ischemic attacks | Mild neurologic deficit with or without imaging confirmation | Moderate neurologic deficit with or without imaging confirmation | - | - | - |
| Definition: A disorder characterize | ed by a brief attack (less than 24 h | nours) of cerebral dysfunction of va | ascular origin, with no persistent n | eurological deficit. | |
| Tremor | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by the uncontrolled shaking mo | evement of the whole body or indiv | ridual parts. | | |
| Trigeminal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by involvement of the trigemina | l nerve (fifth cranial nerve). | | | |
| Vagus nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by involvement of the vagus ne | rve (tenth cranial nerve). | | | ' |
| Vasovagal reaction | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize increase in the stimulation of the | , , , | pressure, bradycardia, and periph | eral vasodilation that may lead to l | oss of consciousness. It results fro | om an |
| Nervous system disorders - | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| Other, specify | symptoms; clinical or diagnostic observations only; intervention not indicated | noninvasive intervention indicated; limiting age-appropriate instrumental ADL | but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | urgent intervention indicated | |
| | | | disabling; limiting self care ADL | | |

| | Pregna | ancy, puerperium and pe | rinatal conditions | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Fetal death | - | | - | - | Fetal loss at |
| | | | | | any |
| | | | | | gestational |
| | | | | | age |
| Definition: A disorder characteriz | ed by death in utero; failure of the | product of conception to show ev | idence of respiration, heartbeat, or | definite movement of a voluntary | muscle after |
| expulsion from the uterus, withou | ut possibility of resuscitation. | | | | |
| Fetal growth retardation | _ | <10% percentile of weight for | <5% percentile of weight for | <1% percentile of weight for | - |
| 9 | | gestational age | gestational age | gestational age | |
| Definition: A disorder characteriz | ed by inhibition of fetal growth resi | ulting in the inability of the fetus to | achieve its potential weight. | ' | , |
| Premature delivery | Delivery of a liveborn infant at | Delivery of a liveborn infant at | Delivery of a liveborn infant at | Delivery of a liveborn infant at | - |
| • | >34 to 37 weeks gestation | >28 to 34 weeks gestation | 24 to 28 weeks gestation | 24 weeks of gestation or less | |
| Definition: A disorder characteriz | ed by delivery of a viable infant be | fore the normal end of gestation. | Typically, viability is achievable be | tween the twentieth and thirty-sev | enth week of |
| gestation. | | · · | | • | |
| Unintended pregnancy | - | - | Unintended pregnancy | - | - |
| Definition: A disorder characteriz | ed by an unexpected pregnancy a | t the time of conception. | | • | |
| Pregnancy, puerperium and | Asymptomatic or mild | Moderate, local or noninvasive | Severe or medically significant | Life-threatening consequences; | Death |
| perinatal conditions - Other, | symptoms; clinical or diagnostic | intervention indicated; limiting | but not immediately life- | urgent intervention indicated | |
| specify | observations only; intervention | instrumental ADL | threatening; hospitalization or | | |
| | not indicated | | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| Psychiatric disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | Severe agitation; hospitalization not indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a state of restlessness asso | ciated with unpleasant feelings of | irritability and tension. | | 1 |
| Anorgasmia | Inability to achieve orgasm not adversely affecting relationship | Inability to achieve orgasm adversely affecting relationship | - | - | - |
| Definition: A disorder characte | rized by an inability to achieve orgas | sm. | _ | _ | ı |
| Anxiety | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization not indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder characte stimulus. | rized by apprehension of danger and | d dread accompanied by restlessn | ess, tension, tachycardia, and dys | pnea unattached to a clearly ident | ifiable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a lack of clear and orderly the | nought and behavior. | | | |
| Delayed orgasm | Delay in achieving orgasm not adversely affecting relationship | Delay in achieving orgasm adversely affecting relationship | - | - | - |
| Definition: A disorder characte | rized by sexual dysfunction characte | rized by a delay in climax. | 1 | T | |
| Delirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional state; limiting self care ADL; hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte reversible condition. | rized by the acute and sudden devel | opment of confusion, illusions, mo | ovement changes, inattentiveness, | agitation, and hallucinations. Usu | ally, it is a |
| Delusions | - | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | rized by false personal beliefs held o | ।<br>contrary to reality, despite contradi | ।<br>ctorv evidence and common sense | 1 - | l |
| Depression | Mild depressive symptoms | Moderate depressive symptoms; limiting instrumental ADL | Severe depressive symptoms;<br>limiting self care ADL;<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; hospitalization indicated | Death |
| Definition: A disorder characte | rized by melancholic feelings of griet | or unhappiness. | | _ | |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., hypomania) | - | - |
| Definition: A disorder characte | rized by an exaggerated feeling of w | ell-being which is disproportionate | to events and stimuli. | | 1 |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; hospitalization indicated | Death |
| Definition: A disorder characte | rized by a false sensory perception i | n the absence of an external stimu | ılus. | • | , |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling asleep, staying asleep or waking up early | Severe difficulty in falling asleep, staying asleep or waking up early | - | - |
| Definition: A disorder characte | rized by difficulty in falling asleep an | d/or remaining asleep. | T | T | 1 |
| Libido decreased | Decrease in sexual interest not adversely affecting relationship | Decrease in sexual interest adversely affecting relationship | - | - | - |
| Definition: A disorder characte | rized by a decrease in sexual desire | T | T | T | 1 |
| Libido increased | Mild increase in sexual interest not adversely affecting relationship | Moderate increase in sexual interest adversely affecting relationship | Severe increase in sexual interest leading to dangerous behavior | - | - |
| Definition: A disorder characte | rized by an increase in sexual desire | ). | | | |
| Mania | Mild manic symptoms (e.g.,<br>elevated mood, rapid thoughts,<br>rapid speech, decreased need<br>for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g.,<br>hypomania; major sexual or<br>financial indiscretions);<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | rized by excitement of psychotic pro | portions manifested by mental and | physical hyperactivity, disorganiz | ation of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |

| | | Psychiatric disord | ders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | ed by a conspicuous change in a p | person's behavior and thinking. | | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(e.g., disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(e.g., paranoid; extreme<br>disorganization); hospitalization<br>not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characterize tumor. | ed by personality change, impaired | d functioning, and loss of touch wi | th reality. It may be a manifestatio | n of schizophrenia, bipolar disorde | er or brain |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an inability to rest, relax or b | pe still. | | | |
| Suicidal ideation | Increased thoughts of death but no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide without serious intent to die which may not require hospitalization | Specific plan to commit suicide with serious intent to die which requires hospitalization | - |
| Definition: A disorder characterize | ed by thoughts of taking one's owr | n life. | | | |
| Suicide attempt | - | - | Suicide attempt or gesture without intent to die which may not require hospitalization | Suicide attempt with intent to die which requires hospitalization | Death |
| Definition: A disorder characterize | ed by self-inflicted harm in an atte | mpt to end one's own life. | | | |
| Psychiatric disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting<br>self care ADL | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |

| | | Renal and urinary dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute kidney injury | mg/dL; creatinine 1.5 - 2.0 x above baseline | Creatinine 2 - 3 x above baseline | Creatinine >3 x baseline or >4.0 mg/dL; hospitalization indicated | Life-threatening consequences; dialysis indicated | Death |
| Definition: A disorder characterize causes (ureteral or bladder outflo | = | on and is traditionally classified a | s pre-renal (low blood flow into kid | ney), renal (kidney damage) and p | oost-renal |
| Bladder perforation | - | Extraperitoneal perforation, indwelling catheter indicated | Intraperitoneal perforation;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by a rupture in the bladder wall | | T | ı | 1 |
| Bladder spasm | Intervention not indicated | Antispasmodics indicated | Hospitalization indicated | - | - |
| Definition: A disorder characterize | ed by a sudden and involuntary co | intraction of the bladder wall. | | | |
| Chronic kidney disease | eGFR (estimated Glomerular<br>Filtration Rate) or CrCl<br>(creatinine clearance) <lln -="" 60<br="">ml/min/1.73 m2 or proteinuria<br/>2+ present; urine<br/>protein/creatinine &gt;0.5</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated | Death |
| Definition: A disorder characterize | ed by gradual and usually perman | ent loss of kidney function resultin | ng in renal failure. | Т | |
| Cystitis noninfective | Microscopic hematuria; minimal increase in frequency, urgency, dysuria, or nocturia; new onset of incontinence | Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characterize | ।<br>ed by inflammation of the bladder। | l | n of the urinary tract. | I | l |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characterize | ed by laboratory test results that ir | dicate blood in the urine. | | | |
| Hemoglobinuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characterize | ed by laboratory test results that in | dicate the presence of free hemo | globin in the urine. | | |
| Proteinuria | 1+ proteinuria; urinary protein<br><1.0 g/24 hrs | Adults: 2+ proteinuria; urinary<br>protein 1.0 - 3.4 g/24 hrs;<br>Pediatric: urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | Adults: urinary protein >=3.5 g/24 hrs;<br>Pediatric: urine P/C >1.9 | - | - |
| Definition: A disorder characterize | ed by laboratory test results that ir | dicate the presence of excessive | protein in the urine. It is predomin | antly albumin, but also globulin. | |
| Renal calculi | Asymptomatic or mild symptoms; occasional use of nonprescription analgesics indicated | Symptomatic; oral antiemetics indicated; around the clock nonprescription analgesics or any oral narcotic analgesics indicated | Hospitalization indicated; IV intervention (e.g., analgesics, antiemetics); elective endoscopic or radiologic intervention indicated | Life-threatening consequences; urgent radiologic, endoscopic or operative intervention indicated | Death |
| Definition: A disorder characterize | ed by the formation of crystals in the | ne pelvis of the kidney. | T | T | T |
| Renal colic | Mild pain not interfering with activity; nonprescription medication indicated | Moderate pain; limiting instrumental ADL; prescription medication indicated | Hospitalization indicated;<br>limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by paroxysmal and severe flant | k marked discomfort radiating to the | ne inguinal area. Often, the cause | is the passage of kidney stones. | |

| Renal and urinary disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Renal hemorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit monitoring indicated | Transfusion, radiation, or<br>hospitalization indicated;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the kidney. | T | 1 | T | |
| Urinary fistula | - | Noninvasive intervention indicated; urinary or suprapubic catheter placement indicated | Limiting self care ADL; elective radiologic, endoscopic or operative intervention indicated; permanent urinary diversion indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between any part of the urinary | system and another organ or anato | omic site. | |
| Urinary frequency | Present rized by urination at short intervals. | Limiting instrumental ADL; medical management indicated | - | - | - |
| | | Spontaneous: pade indicated: | Intervention indicated (a.g. | | |
| Urinary incontinence | Occasional (e.g., with coughing, sneezing, etc.), pads not indicated | Spontaneous; pads indicated;<br>limiting instrumental ADL | Intervention indicated (e.g., clamp, collagen injections); operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder character | rized by inability to control the flow o | f urine from the bladder. | | | |
| Urinary retention | Urinary, suprapubic or intermittent catheter placement not indicated; able to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective operative or radiologic intervention indicated; substantial loss of affected kidney function or mass | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by accumulation of urine within | the bladder because of the inabil | ity to urinate. | , | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ function (e.g., hydronephrosis, or renal dysfunction); elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by blockage of the normal flow | of contents of the urinary tract. | | | |
| Urinary tract pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the urinary tract. | ı | T | |
| Urinary urgency | Present | Limiting instrumental ADL; medical management indicated | - | - | - |
| Definition: A disorder character | rized by a sudden compelling urge to | urinate. | 1 | 1 | |
| Urine discoloration | Present | - | - | - | - |
| Definition: A disorder character | rized by a change in the color of the | urine. | | | |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Rep | productive system and bi | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Azoospermia | - | - | Absence of sperm in ejaculate | - | - |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate complete absence of sperr | natozoa in the semen. | <u> </u> | |
| Breast atrophy | Minimal asymmetry; minimal atrophy | Moderate asymmetry; moderate atrophy | Asymmetry >1/3 of breast volume; severe atrophy | - | - |
| Definition: A disorder characteriz | ed by underdevelopment of the bro | east. | | | |
| Breast pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the breast region. | | | |
| Dysmenorrhea | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by abnormally painful abdomina | al cramps during menses. | _ | _ | |
| Dyspareunia | Mild discomfort or pain<br>associated with vaginal<br>penetration; discomfort relieved<br>with use of vaginal lubricants or<br>estrogen | Moderate discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>partially relieved with use of<br>vaginal lubricants or estrogen | Severe discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>unrelieved by vaginal lubricants<br>or estrogen | - | - |
| Definition: A disorder characteriz | ed by painful or difficult coitus. | , | , | ' | ı |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde ejaculation | - | - | - |
| Definition: A disorder characteriz | '<br>ed by problems related to ejaculat | ion. This category includes prema | '<br>ture, delayed, retrograde and pair | ful ejaculation. | 1 |
| Erectile dysfunction | Decrease in erectile function<br>(frequency or rigidity of<br>erections) but intervention not<br>indicated (e.g., medication or<br>use of mechanical device,<br>penile pump) | Decrease in erectile function<br>(frequency/rigidity of erections),<br>erectile intervention indicated,<br>(e.g., medication or mechanical<br>devices such as penile pump) | Decrease in erectile function (frequency/rigidity of erections) but erectile intervention not helpful (e.g., medication or mechanical devices such as penile pump); placement of a permanent penile prosthesis indicated (not previously present) | - | - |
| Definition: A disorder characteriz | ed by the persistent or recurrent in | nability to achieve or to maintain a | n erection during sexual activity. | | ' |
| Fallopian tube obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the contents in the fallopian tub | e. | T | T |
| Fallopian tube stenosis | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| | ed by a narrowing of the fallopian | tube lumen. | Ι | T | |
| Female genital tract fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an abnormal communication | | ystem organ and another organ o | r anatomic site. | |
| Feminization acquired | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by the development of seconda | ary female sex characteristics in m | ales due to extrinsic factors. | T | I |
| Genital edema | Mild swelling or obscuration of anatomic architecture on close inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour | Lymphorrhea; gross deviation<br>from normal anatomic contour;<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by swelling due to an excessive | e accumulation of fluid in the genit | als. | Γ | |
| Gynecomastia | Asymptomatic breast enlargement | Symptomatic (e.g., pain or psychosocial impact) | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by excessive development of the | ne breasts in males. | | | |
| Hematosalpinx | Minimal bleeding identified on imaging study or laparoscopy; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | zed by the presence of blood in a fa | allopian tube. | T | T | 1 |
| Irregular menstruation | Intermittent menses with skipped menses for no more than 1 to 3 months | Intermittent menses with skipped menses for more than 4 to 6 months | Persistent amenorrhea for more than 6 months | - | - |
| Definition: A disorder characterization | zed by irregular cycle or duration of | menses. | | | |
| Lactation disorder | Mild changes in lactation, not significantly affecting production or expression of breast milk | Changes in lactation,<br>significantly affecting breast<br>production or expression of<br>breast milk | - | - | - |
| Definition: A disorder characterize | zed by disturbances of milk secretion | on. It is not necessarily related to p | pregnancy that is observed in fema | ales and can be observed in males | 3.<br>T |
| Menorrhagia | Mild; iron supplements indicated | Moderate symptoms; medical intervention indicated (e.g., hormones) | Severe; transfusion indicated;<br>surgical intervention indicated<br>(e.g., hysterectomy) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterization | zed by abnormally heavy vaginal bl | eeding during menses. | | | |
| Nipple deformity | Asymptomatic; asymmetry with slight retraction and/or thickening of the nipple areolar complex | Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex | - | - | - |
| Definition: A disorder characterization | zed by a malformation of the nipple | | | | |
| Oligospermia | Sperm concentration >48 million/mL or motility >68% | Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Sperm concentration <13 million/mL or motility <32% | - | - |
| Definition: A disorder characteriz | zed by a decrease in the number of | spermatozoa in the semen. | | | |
| Ovarian hemorrhage | Minimal bleeding identified on imaging study or laproscopy; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterization | zed by bleeding from the ovary. | | | | |
| Ovarian rupture | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterization | '<br>zed by tearing or disruption of the o | varian tissue. | • | ' | ı |
| Ovulation pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterizovarian follicle. | zed by marked discomfort sensation | , | | time of the discharge of the ovum | from the |
| Pelvic floor muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic, not interfering with bladder, bowel, or vaginal function; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterization | zed by a reduction in the strength o | f the muscles of the pelvic floor. | | | |
| Pelvic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterization | zed by marked discomfort sensation | n in the pelvis. | | | |
| Penile pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterization | zed by marked discomfort sensation | n in the penis. | | | |
| Perineal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterization | zed by a sensation of marked disco | mfort in the area between the ger | nital organs and the anus. | | |
| Premature menopause | - | - | Present | - | - |
| • | ा<br>zed by ovarian failure before the ag | i<br>le of 40. Symptoms include hot fla | 1 | and a decrease in sex drive | I |
| Prostatic hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by bleeding from the prostate of | gland. | | | |
| Prostatic obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by compression of the urethra | secondary to enlargement of the p | '<br>rostate gland. This results in voidi | ng difficulties (straining to void, slo | ow urine |
| stream, and incomplete emptying | of the bladder). | | | | |
| Prostatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the prostate gland. | ı | • | 1 |
| Scrotal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ।<br>ed by marked discomfort sensatio | 1 | I | l | I |
| Spermatic cord hemorrhage | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| opormulae cord nomermage | imaging study; intervention not indicated | intervention indicated | indicated; radiologic or endoscopic intervention | urgent operative intervention indicated | Dodui |
| Definition. A discardes absorbesis | | - and | indicated | | |
| | ed by bleeding from the spermatic | | Covers summataness along | | |
| Spermatic cord obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the contents of the spermatic c | ord. | | 1 |
| Testicular disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic but not interfering with urination or sexual activities; intervention not indicated; limiting instrumental ADL | Severe symptoms; interfering with urination or sexual function; limiting self care ADL; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the testis. | | | | |
| Testicular hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the testis. | | _ | | |
| Testicular pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the testis. | | | |
| Uterine fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the uterus and another | organ or anatomic site. | • | , |
| Uterine hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the uterus. | 1 | <b>.</b> | | 1 |
| Uterine obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by blockage of the uterine outle | et. | | | |
| Uterine pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the uterus. | • | • | |
| Vaginal discharge | Mild vaginal discharge (greater than baseline for patient) | Moderate to heavy vaginal discharge; use of perineal pad or tampon indicated | - | - | - |
| Definition: A disorder characterize | i<br>ed by vaginal secretions. Mucus n | 1 | I<br>discharged from the vagina natura | ı<br>Ily, especially during the childhear | ing years. |
| Vaginal dryness | Mild vaginal dryness not interfering with sexual function | Moderate vaginal dryness interfering with sexual function or causing frequent discomfort | Severe vaginal dryness resulting in dyspareunia or severe discomfort | - | - |
| Definition: A disorder characterize | ed by an uncomfortable feeling of | itching and burning in the vagina. | | | |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Vaginal fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterization | zed by an abnormal communication | between the vagina and another | organ or anatomic site. | | |
| Vaginal hemorrhage | Minimal bleeding identified on clinical exam or imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteria | zed by bleeding from the vagina. | | | | |
| Vaginal inflammation | Mild discomfort or pain, edema, or redness | Moderate discomfort or pain, edema, or redness; limiting instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal<br>ulceration; life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteria | zed by inflammation involving the v | agina. Symptoms may include red | dness, edema, marked discomfort | and an increase in vaginal dischar | ge. |
| Vaginal obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteria | zed by blockage of vaginal canal. | | | | |
| √aginal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteria | zed by a sensation of marked disco | omfort in the vagina. | | | |
| Vaginal perforation | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a rupture in the vaginal wall. | | | | |
| Vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or<br>shortening not interfering with<br>physical examination | Vaginal narrowing and/or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | - | Death |
| Definition: A disorder characteria | zed by a narrowing of the vaginal c | anal. | • | ' | • |
| Vaginismus | Mild discomfort or pain<br>associated with vaginal<br>spasm/tightening; no impact<br>upon sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spasm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal<br>spasm/tightening; unable to<br>tolerate vaginal penetration or<br>physical examination | - | - |
| Definition: A disorder characterizintercourse. | zed by involuntary spasms of the po | elvic floor muscles, resulting in pa | thologic tightness of the vaginal w | all during penetration such as duri | ng sexua |
| Reproductive system and breas<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adult respiratory distress | • | | Present with radiologic findings; | Life-threatening respiratory or | Death |
| syndrome | | | intubation not indicated | hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte<br>surgery. | erized by progressive and life-threater | ning pulmonary distress in the abs | ence of an underlying pulmonary | condition, usually following major t | rauma o |
| Allergic rhinitis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| | erized by an inflammation of the nasal | | = : | = | ay also |
| | es of the sinuses, eyes, middle ear, a | ind pharynx. Symptoms include sr | 1 | | |
| Apnea | - | - | Present; medical intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | erized by cessation of breathing. | | | 1 | I |
| Aspiration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Altered eating habits; coughing or choking episodes after eating or swallowing; medical intervention indicated (e.g., suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); hospitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | erized by inhalation of solids or liquids | s into the lungs. | _ | | |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | erized by the collapse of part or the er | _ | | | - · |
| Bronchial fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL; endoscopic or operative intervention indicated (e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild wheezing); endoscopic evaluation indicated; radiographic evidence of atelectasis/lobar collapse; medical management indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | erized by blockage of a bronchus pass | sage, most often by bronchial sec | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the bronchial | tube. | T | ı | |
| Bronchopleural fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL; endoscopic or operative intervention indicated (e.g., stent or primary closure) | Life-threatening consequences; urgent operative intervention with thoracoplasty, chronic open drainage or multiple thoracotomies indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between a bronchus and the plei | ural cavity. | | |
| Bronchopulmonary hemorrha | ge Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic, endoscopic, or operative intervention indicated (e.g., | Life-threatening respiratory or hemodynamic compromise; intubation or urgent intervention | Death |

| | Respiratory, thoracic and mediastinal disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bronchospasm Definition: A disorder characterize | Mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL smooth muscles of the bronchial v | Limiting self care ADL; oxygen saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Chylothorax | Asymptomatic; clinical or | Symptomatic; thoracentesis or | | Life threatening requirators or | Death |
| Chylotholax | diagnostic observations only;<br>intervention not indicated | tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Deam |
| Definition: A disorder characterize | ed by milky pleural effusion (abnor | rmal collection of fluid) resulting fro | om accumulation of lymph fluid in | the pleural cavity. | |
| Cough | Mild symptoms; nonprescription intervention indicated | Moderate symptoms, medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize by a distinctive sound. | ed by sudden, often repetitive, spa | asmodic contraction of the thoracion | c cavity, resulting in violent release | e of air from the lungs and usually a | accompanied |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with minimal exertion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an uncomfortable sensation | of difficulty breathing. | 1 | T | T |
| Epistaxis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated (e.g., nasal packing, cauterization; topical vasoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the nose. | | T | T | ı |
| Hiccups | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe symptoms; interfering with sleep; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by repeated gulp sounds that re | esult from an involuntary opening | and closing of the glottis. This is a | ttributed to a spasm of the diaphra | igm. |
| Hoarseness | Mild or intermittent voice<br>change; fully understandable;<br>self-resolves | Moderate or persistent voice changes; may require occasional repetition but understandable on telephone; medical evaluation indicated | Severe voice changes including predominantly whispered speech | - | - |
| Definition: A disorder characterize | ed by harsh and raspy voice arisir | ng from or spreading to the larynx. | T | T | T |
| Hypoxia Definition: A disorder characterizate in the second control of the second contr | -<br>ed by a decrease in the level of ox | Decreased oxygen saturation with exercise (e.g., pulse oximeter <88%); intermittent supplemental oxygen in the body | Decreased oxygen saturation at<br>rest (e.g., pulse oximeter <88%<br>or PaO2 <=55 mm Hg) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Laryngeal edema | Asymptomatic; clinical or | Symptomatic; medical | Stridor; respiratory distress; | Life-threatening airway | Death |
| au yr gan acomu | diagnostic observations only;<br>intervention not indicated | intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | hospitalization indicated | compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Joan |
| Definition: A disorder characterize | ed by swelling due to an excessive | e accumulation of fluid in the laryn | X. | Ι | |
| Laryngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characterize | ed by an abnormal communication | between the larynx and another | organ or anatomic site. | | |
| Laryngeal hemorrhage | Mild cough or trace hemoptysis;<br>laryngoscopic findings | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characterize | ed by bleeding from the larynx. | | Τ | Γ | |
| Laryngeal inflammation | Mild sore throat; raspy voice | Moderate sore throat; analgesics indicated | Severe throat pain; endoscopic intervention indicated | - | - |
| Definition: A disorder characterize | ed by an inflammation involving th | e larynx. | | | |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngeal mucositis Definition: A disorder characterize | Endoscopic findings only; mild discomfort with normal intake | Moderate discomfort; altered oral intake | Severe pain; severely altered eating/swallowing; medical intervention indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | 1 | | | I | <b>5</b> " |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by blockage of the laryngeal air | rway. | | | |
| Laryngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a narrowing of the laryngeal | airway. | | | |
| Laryngopharyngeal dysesthesia | Mild symptoms; no anxiety; intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspnea and swallowing difficulty; limiting self care ADL | Life-threatening consequences | Death |
| Definition: A disorder characterize | ed by an uncomfortable persistent | sensation in the area of the laryn | gopharynx. | | |
| Laryngospasm | - | Transient episode; intervention not indicated | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| Definition: A disorder characterize | ed by paroxysmal spasmodic mus | cular contraction of the vocal cord | S. | | |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated<br>(e.g., hemostasis of bleeding<br>site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the mediastin | um. | | | |
| Nasal congestion | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Associated with bloody nasal discharge or epistaxis | - | - |
| Definition: A disorder characterize | ed by obstruction of the nasal pas | sage due to mucosal edema. | | | |
| Pharyngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | n between the pharynx and anothe | er organ or anatomic site. | | |
| Pharyngeal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | ed by bleeding from the pharynx. | | | | |
| Pharyngeal mucositis | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics indicated; altered oral intake; limiting instrumental ADL | Severe pain; unable to<br>adequately aliment or hydrate<br>orally; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an inflammation involving th | e mucous membrane of the phary | rnx. | | |
| Pharyngeal necrosis | - | - | Inability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | <u> </u> |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | zed by a necrotic process occurring | | | | |
| Pharyngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characteriz | zed by a narrowing of the pharynge | al airway. | | | |
| Pharyngolaryngeal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by marked discomfort sensation | n in the pharyngolaryngeal region. | 1 | I | ı |
| Pleural effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., diuretics or limited therapeutic thoracentesis) | Symptomatic with respiratory distress and hypoxia; surgical intervention including chest tube or pleurodesis indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | zed by an increase in amounts of flo | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomfo | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage confirmed by thoracentesis | Symptomatic or associated with pneumothorax; chest tube drainage indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the pleural ca | vity. | | | |
| Pleuritic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by marked discomfort sensation | n in the pleura. | | | |
| Pneumonitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; oxygen indicated | Life-threatening respiratory compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characterize | zed by inflammation focally or diffus | sely affecting the lung parenchyma | a. | Т | I |
| Pneumothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., tube placement without sclerosis) | Sclerosis and/or operative intervention indicated; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by abnormal presence of air in | the pleural cavity resulting in the o | collapse of the lung. | | |
| Postnasal drip | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | zed by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | |
| Productive cough | Occasional/minimal production of sputum with cough | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | - | - |
| | zed by expectorated secretions upo | | Covere duannes en duannes | Life threatening rearists | Dooth |
| Pulmonary edema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspnea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspnea or dyspnea at rest; oxygen indicated; limiting self care ADL | Life-threatening respiratory<br>compromise; urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder characterize | zed by accumulation of fluid in the I | ung tissues that causes a disturba | ince of the gas exchange that may | / lead to respiratory failure. | |
| Pulmonary fibrosis | Mild hypoxemia; radiologic pulmonary fibrosis <25% of lung volume | radiographic pulmonary fibrosis<br>25 - 50% | right-sided heart failure;<br>radiographic pulmonary fibrosis<br>>50 - 75% | Life-threatening consequences (e.g., hemodynamic/pulmonary complications); intubation with ventilatory support indicated; radiographic pulmonary fibrosis >75% with severe honeycombing | Death |
| Definition: A disorder characterize | zed by the replacement of the lung | tissue by connective tissue, leadir | ng to progressive dyspnea, respira | tory failure or right heart failure. | ı |
| Pulmonary fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Limiting self care ADL;<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | Grade 3 | 4 | 5 |
| | | | | 4 | 5 |
| Pulmonary hypertension | Minimal dyspnea; findings on physical exam or other evaluation | Moderate dyspnea, cough;<br>requiring evaluation by cardiac<br>catheterization and medical<br>intervention | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening airway<br>consequences; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| Definition: A disorder characteriz | ed by an increase in pressure with | in the pulmonary circulation due to | lung or heart disorder. | | |
| Respiratory failure | - | - | - | Life-threatening consequences; urgent intervention, intubation, or ventilatory support indicated | Death |
| Definition: A disorder characteriz<br>with an increase in arterial levels | ed by impaired gas exchange by the of carbon dioxide. | he respiratory system resulting in | nypoxemia and a decrease in oxy | genation of the tissues that may be | e associate |
| Retinoic acid syndrome | Fluid retention; <3 kg of weight gain; intervention with fluid restriction and/or diuretics indicated | Moderate signs or symptoms; steroids indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; ventilatory support indicated | Death |
| Definition: A disorder characteriz retinoic acid. | ed by weight gain, dyspnea, pleura | al and pericardial effusions, leukoo | cytosis and/or renal failure original | ly described in patients treated wit | h all-trans |
| Sinus disorder | Asymptomatic mucosal crusting; blood-tinged secretions | Symptomatic stenosis or edema/narrowing interfering with airflow; limiting instrumental ADL | Stenosis with significant nasal obstruction; limiting self care ADL | Necrosis of soft tissue or bone; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the paranasa | al sinuses. | | | |
| Sleep apnea | Snoring and nocturnal sleep arousal without apneic periods | Moderate apnea and oxygen<br>desaturation; excessive daytime<br>sleepiness; medical evaluation<br>indicated; limiting instrumental<br>ADL | Oxygen desaturation;<br>associated with hypertension;<br>medical intervention indicated;<br>limiting self care ADL | Cardiovascular or<br>neuropsychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by cessation of breathing for sh | ı | ı | I | ı |
| Sneezing | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | red by the involuntary expulsion of | air from the nose. | <u> </u> | Г | 1 |
| Sore throat | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to swallow | - | - |
| Definition: A disorder characteriz | ed by of marked discomfort in the | throat | | | |
| Stridor | - | - | Respiratory distress limiting self care ADL; medical intervention indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | red by a high pitched breathing sou | 1 | r e | | |
| Tracheal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the trachea and another | organ or anatomic site. | | |
| Tracheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe pain; hemorrhage or respiratory symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an inflammation involving the | | | | |
| Tracheal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Stridor or respiratory distress<br>limiting self care ADL;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | · | i ' | İ | i | 1 |

| , | | | | Respiratory, thoracic and mediastinal disorders |
|---|---|---|---|---|
| | | Grade | | |
| 1 | 2 | 3 | 4 | 5 |
| Mild or intermittent change from normal voice | Moderate or persistent change from normal voice; still understandable | Severe voice changes including predominantly whispered speech; may require frequent repetition or face-to-face contact for understandability; may | - | - |
| led by a change in the sound and/o | l<br>or speed of the voice. | require assistive technology | | |
| Detectable airway noise with minimal symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe respiratory symptoms<br>limiting self care ADL; oxygen<br>therapy or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| ed by a high-pitched, whistling sou | ind during breathing. It results fror | n the narrowing or obstruction of the | ne respiratory airways. | |
| Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| 9 | normal voice ad by a change in the sound and/or Detectable airway noise with minimal symptoms ad by a high-pitched, whistling sou Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | from normal voice; still understandable ad by a change in the sound and/or speed of the voice. Detectable airway noise with minimal symptoms Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention indicated; limiting instrumental ADL Moderate; minimal, local or noninvasive intervention indicated; limiting age- | from normal voice from normal voice; still understandable predominantly whispered speech; may require frequent repetition or face-to-face contact for understandability; may require assistive technology red by a change in the sound and/or speed of the voice. Detectable airway noise with minimal symptoms Moderate symptoms; medical intervention indicated; limiting instrumental ADL Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated which indicated symptoms to mild symptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; limiting age-appropriate instrumental ADL prolongation of existing | normal voice from normal voice; still understandable speech; may require frequent repetition or face-to-face contact for understandability; may require assistive technology. In the sound and/or speed of the voice. Detectable airway noise with minimal symptoms intervention indicated; limiting instrumental ADL In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated indicated. In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated. In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated. In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated. In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated. In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated. In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated. In the sound and/or speed of the voice. Severe respiratory symptoms limiting self care ADL; oxygen therapy or hospitalization indicated. In the sound and/or speed of the voice. Severe respiratory symptoms. In the sound and/or speed of the voice. Severe respiratory symptoms. In the sound and/or speed of the voice. Severe respiratory symptoms. In the sound and/or speed of the voice. Severe respiratory symptoms limiting aperate and |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | Grade 3 | 4 | 5 |
| Alopecia | Hair loss of <50% of normal for | Hair loss of >=50% normal for | J | 4 | 3 |
| Alopecia | that individual that is not | that individual that is readily | - | - | - |
| | obvious from a distance but only | apparent to others; a wig or hair | | | |
| | on close inspection; a different | piece is necessary if the patient | | | |
| | hair style may be required to | desires to completely | | | |
| | cover the hair loss but it does | camouflage the hair loss; | | | |
| | not require a wig or hair piece to | associated with psychosocial | | | |
| | camouflage | impact | | | |
| Definition: Δ disorder character | ized by a decrease in density of hair | | l<br>ndividual at a given age and hody | location | |
| | | · | | location. | |
| Body odor | Mild odor; physician intervention | Pronounced odor; psychosocial | - | - | - |
| | not indicated; self care | impact; patient seeks medical | | | |
| | interventions | intervention | | | |
| Definition: A disorder character | ized by an abnormal body smell res | ulting from the growth of bacteria | on the body. | 1 | 1 |
| Bullous dermatitis | Asymptomatic; blisters covering | Blisters covering 10 - 30% BSA; | Blisters covering >30% BSA; | Blisters covering >30% BSA; | Death |
| | <10% BSA | painful blisters; limiting | limiting self care ADL | associated with fluid or | |
| | | instrumental ADL | | electrolyte abnormalities; ICU | |
| | | | | care or burn unit indicated | |
| Definition: A disorder character | ized by inflammation of the skin cha | racterized by the presence of bull | ae which are filled with fluid. | | |
| Ory skin | Covering <10% BSA and no | Covering 10 - 30% BSA and | Covering >30% BSA and | _ | _ |
| 2., c | associated erythema or pruritus | associated with erythema or | associated with pruritus; limiting | | |
| | according of prantac | pruritus; limiting instrumental | self care ADL | | |
| | | ADL | Son Gare 7 (SE | | |
| Definition: A disorder character | ized by flaky and dull skin; the peres | 1 | a nanony thin toyture | ! | ļ |
| | ized by flaky and dull skin; the pores | _ · | 1 | | |
| Erythema multiforme | Target lesions covering <10% | Target lesions covering 10 - | Target lesions covering >30% | Target lesions covering >30% | Death |
| | BSA and not associated with | 30% BSA and associated with | BSA and associated with oral or | BSA; associated with fluid or | |
| | skin tenderness | skin tenderness | genital erosions | electrolyte abnormalities; ICU | |
| | | | | care or burn unit indicated | |
| Definition: A disorder character | ized by target lesions (a pink-red rin | g around a pale center). | | _ | _ |
| Erythroderma | - | Erythema covering >90% BSA | Erythema covering >90% BSA | Erythema covering >90% BSA | Death |
| | | without associated symptoms; | with associated symptoms (e.g., | with associated fluid or | |
| | | limiting instrumental ADL | pruritus or tenderness); limiting | electrolyte abnormalities; ICU | |
| | | | self care ADL | care or burn unit indicated | |
| Definition: A disorder character | ized by generalized inflammatory er | vthema and exfoliation. The inflan | nmatory process involves > 90% c | of the body surface area. | ' |
| Fat atrophy | Covering <10% BSA and | Covering 10 - 30% BSA and | Covering >30% BSA; | 1_ | |
| at all opiny | | | | | - |
| | asymptomatic | associated with erythema or tenderness; limiting instrumental | associated with erythema or | | |
| | | ADL | ADL | | |
| Saffattian Autorologists | | /\DL | I NOL | I | 1 |
| | ized by shrinking of adipose tissue. | | | | |
| Hirsutism | In women, increase in length, | In women, increase in length, | - | - | - |
| | thickness or density of hair in a | thickness or density of hair in a | | | |
| | male distribution that the patient | male distribution that requires | | | |
| | is able to camouflage by | daily shaving or consistent | | | |
| | periodic shaving, bleaching, or | destructive means of hair | | | |
| | removal of hair | removal to camouflage; | | | |
| | | associated with psychosocial | | | |
| | | impact | | | |
| | ized by the presence of excess hair | growth in women in anatomic site | s where growth is considered to b | e a secondary male characteristic | and unde |
| androgen control (beard, mous | tache, chest, abdomen) | Г | T | 1 | |
| Hyperhidrosis | Limited to one site (palms, | Involving >1 site; patient seeks | Generalized involving sites | - | - |
| | soles, or axillae); self care | medical intervention; associated | other than palms, soles, or | | |
| | interventions | with psychosocial impact | axillae; associated with | | |
| | | | electrolyte/hemodynamic | | |
| | | | imbalance | | |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal | Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair | - | - | - |
| Definition: A disorder characterize | ad by bair density or length beyond | removal to camouflage;<br>associated with psychosocial<br>impact | a particular body region, for a part | icular ago or raco | |
| | ed by fiall defisity of length beyon | | a particular body region, for a part | | <b>.</b> |
| Hypohidrosis Definition: A disorder characterize | ed by reduced sweating. | Symptomatic; limiting instrumental ADL | Increase in body temperature;<br>limiting self care ADL | Heat stroke | Death |
| Lipohypertrophy | Asymptomatic and covering <10% BSA | Covering 10 - 30% BSA and associated tenderness; limiting instrumental ADL | Covering >30% BSA and<br>associated tenderness and<br>narcotics or NSAIDs indicated;<br>lipohypertrophy; limiting self<br>care ADL | - | - |
| Definition: A disorder characterize | ed by hypertrophy of the subcutan | eous adipose tissue at the site of | nultiple subcutaneous injections o | of insulin. | ļ |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characterize | ed by a change in the color of the | nail plate. | | | |
| Nail loss | Asymptomatic separation of the nail bed from the nail plate or nail loss | Symptomatic separation of the nail bed from the nail plate or nail loss; limiting instrumental ADL | - | - | - |
| Definition: A disorder characterize | ed by loss of all or a portion of the | nail. | | | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characterize | ed by vertical or horizontal ridges | on the nails. | | | |
| Pain of skin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort sensation | n in the skin. | <b>.</b> | 1 | 1 |
| Palmar-plantar erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling,<br>blisters, bleeding, edema, or<br>hyperkeratosis) with pain;<br>limiting instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>edema, or hyperkeratosis) with<br>pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by redness, marked discomfort | , swelling, and tingling in the palm | s of the hands or the soles of the | feet. | 1 |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated | - | - |
| Definition: A disorder characterize | ed by swelling due to an excessive | accumulation of fluid around the | orbits of the face. | | |
| Photosensitivity | Painless erythema and erythema covering <10% BSA | Tender erythema covering 10 -<br>30% BSA | Erythema covering >30% BSA and erythema with blistering; photosensitivity; oral corticosteroid therapy indicated; pain control indicated (e.g., narcotics or NSAIDs) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an increase in sensitivity of t | he skin to light. | | | |

| | Skin and subcutaneous tissue disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical intervention indicated | Intense or widespread;<br>intermittent; skin changes from<br>scratching (e.g., edema,<br>papulation, excoriations,<br>lichenification, oozing/crusts);<br>oral intervention indicated; | Intense or widespread;<br>constant; limiting self care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | - | - |
| Definition: A disorder characteriz | and by an intense itahing concetion | limiting instrumental ADL | | | |
| Purpura | Combined area of lesions covering <10% BSA | Combined area of lesions covering 10 - 30% BSA; bleeding with trauma | Combined area of lesions covering >30% BSA; spontaneous bleeding | -<br>Nder lesions are usually a darker r | - |
| and eventually become a brownis | | in and mucous membrane. Newer | resions appear reduisir in color. C | older lesions are usually a darker p | ourpie color |
| Rash acneiform | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10 - 30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| Definition: A disorder characteriz | ed by an eruption of papules and p | oustules, typically appearing in fac | e, scalp, upper chest and back. | T | |
| Rash maculo-papular | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness) | Macules/papules covering 10 -<br>30% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness); limiting<br>instrumental ADL | Macules/papules covering >30% BSA with or without associated symptoms; limiting self care ADL | - | - |
| | ed by the presence of macules (flat<br>apper trunk, spreading centripetally | | nown as morbillform rash, it is one | of the most common cutaneous a | dverse |
| Scalp pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the skin covering the top and | the back of the head. | | |
| Skin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA; associated with ulceration | - | - |
| Definition: A disorder characteriz | ed by the degeneration and thinning | | I | | |
| Skin hyperpigmentation | Hyperpigmentation covering <10% BSA; no psychosocial impact | Hyperpigmentation covering >10% BSA; associated psychosocial impact | - | - | - |
| Definition: A disorder characteriz | ed by darkening of the skin due to | excessive melanin deposition. | 1 | | Г |
| Skin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering >10%<br>BSA; associated psychosocial<br>impact | - | - | - |
| Definition: A disorder characteriz | ed by loss of skin pigment. | | | | |
| Skin induration | Mild induration, able to move skin parallel to plane (sliding) and perpendicular to skin (pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration, unable to<br>slide or pinch skin; limiting joint<br>movement or orifice (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| Definition: A disorder characteriz | red by an area of hardness in the s | kin. | I | | Т |
| Skin ulceration | Combined area of ulcers <1 cm;<br>nonblanchable erythema of<br>intact skin with associated<br>warmth or edema | Combined area of ulcers 1 - 2<br>cm; partial thickness skin loss<br>involving skin or subcutaneous<br>fat | Combined area of ulcers >2 cm;<br>full-thickness skin loss involving<br>damage to or necrosis of<br>subcutaneous tissue that may<br>extend down to fascia | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or supporting structures with or without full thickness skin loss | Death |
| Definition: A disorder characteriz | ed by circumscribed, inflammatory | and necrotic erosive lesion on the | e skin. | | |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome | - | - | Skin sloughing covering <10%<br>BSA with associated signs (e.g.,<br>erythema, purpura, epidermal<br>detachment and mucous<br>membrane detachment) | Skin sloughing covering 10 -<br>30% BSA with associated signs<br>(e.g., erythema, purpura,<br>epidermal detachment and<br>mucous membrane<br>detachment) | Death |
| | ed by less than 10% total body ski | n area separation of dermis. The | syndrome is thought to be a hyper | sensitivity complex affecting the sl | kin and the |
| Telangiectasia | Telangiectasias covering <10%<br>BSA | Telangiectasias covering >10%<br>BSA; associated with<br>psychosocial impact | - | - | - |
| | ed by local dilatation of small vess | els resulting in red discoloration o | the skin or mucous membranes. | | |
| Toxic epidermal necrolysis | - | - | - | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| Definition: A disorder characteriz mucous membranes. | ed by greater than 30% total body | skin area separation of dermis. Ti | he syndrome is thought to be a hy | persensitivity complex affecting the | e skin and the |
| Urticaria | Urticarial lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesions covering 10 - 30% BSA; oral intervention indicated | Urticarial lesions covering >30%<br>BSA; IV intervention indicated | - | - |
| Definition: A disorder characteriz | ed by an itchy skin eruption charac | cterized by wheals with pale interior | ors and well-defined red margins. | | |
| Skin and subcutaneous tissue disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Social circumstances | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Menopause | Menopause occurring at age 46 - 53 years of age | Menopause occurring at age 40 - 45 years of age | Menopause occurring before age 40 years of age | - | - |
| Definition: A disorder characteriz | ed by the permanent cessation of | menses, usually defined by 12 cor | nsecutive months of amenorrhea i | n a woman over 45 years of age. | |
| Social circumstances - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| 1 | | | disabling; limiting self care ADL | | |

| Surgical and medical procedures | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Surgical and medical procedures - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Capillary leak syndrome | - | Symptomatic; medical intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by leakage of intravascular fluid | · | | <del>-</del> | |
| leaky capillaries following shock failure. | syndromes, low-flow states, ischei | mia-reperfusion injuries, toxemias, | medications, or poisoning. It can | lead to generalized edema and m | ultiple organ |
| Flushing | Asymptomatic; clinical or diagnostic observations only; | Moderate symptoms; medical intervention indicated; limiting | Symptomatic, associated with hypotension and/or tachycardia; | - | - |
| | intervention not indicated | instrumental ADL | limiting self care ADL | | ļ |
| | zed by episodic reddening of the fa | | | <u> </u> | |
| Hematoma | Mild symptoms; intervention not indicated | Minimally invasive evacuation or aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a localized collection of bloc | od, usually clotted, in an organ, spa | ace, or tissue, due to a break in the | e wall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by an uncomfortable and temper | orary sensation of intense body wa | armth, flushing, sometimes accom | panied by sweating upon cooling. | 1 |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic<br>BP 140 - 159 mm Hg or<br>diastolic BP 90 - 99 mm Hg);<br>medical intervention indicated;<br>recurrent or persistent (>=24<br>hrs); symptomatic increase by | Stage 2 hypertension (systolic BP >=160 mm Hg or diastolic BP >=100 mm Hg); medical intervention indicated; more than one drug or more intensive therapy than previously used | Life-threatening consequences<br>(e.g., malignant hypertension,<br>transient or permanent<br>neurologic deficit, hypertensive<br>crisis); urgent intervention<br>indicated | Death |
| | | >20 mm Hg (diastolic) or to<br>>140/90 mm Hg if previously<br>WNL; monotherapy indicated<br>Pediatric: recurrent or persistent<br>(>=24 hrs) BP >ULN;<br>monotherapy indicated | indicated Pediatric: Same as adult | Pediatric: Same as adult | |
| Definition: A disorder characterize | zed by a pathological increase in bl | lood pressure; a repeatedly elevat | ion in the blood pressure exceedir | ng 140 over 90 mm Hg. | , |
| Hypotension | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention or hospitalization indicated | Life-threatening and urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a blood pressure that is belo | ow the normal expected for an indi | vidual in a given environment. | | |
| Lymph leakage | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | red by the loss of lymph fluid into the | ne surrounding tissue or body cavi | ty. | T | |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery skin texture; papillary formation; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by excessive fluid collection in | tissues that causes swelling. | _ | _ | |
| Lymphocele | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | - | - |
| Definition: A disorder characterized by a cystic lesion containing lymph. | | | | | |
| Peripheral ischemia | - | Brief (<24 hrs) episode of ischemia managed non-surgically and without permanent deficit | Recurring or prolonged (>=24 hrs) and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by impaired circulation to an ex | ktremity. | | | |
| Phlebitis | - | Present | - | - | - |
| Definition: A disorder characteriz | ed by inflammation of the wall of a | vein. | | | |
| Superficial thrombophlebitis | - | Present | - | - | - |
| Definition: A disorder characteriz | zed by a blood clot and inflammatic | on involving a superficial vein of the | e extremities. | | |

| | Vascular disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening consequences;<br>urgent multi-modality<br>intervention indicated (e.g.,<br>lysis, thrombectomy, surgery) | Death |
| Definition: A disorder characterize cough, orthopnea and headache | ed by obstruction of the blood flow | in the superior vena cava. Signs | and symptoms include swelling an | d cyanosis of the face, neck, and | upper arms, |
| Thromboembolic event | Venous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | thrombus), medical intervention | Life-threatening (e.g., pulmonary embolism, cerebrovascular event, arterial insufficiency); hemodynamic or neurologic instability; urgent intervention indicated | Death |
| Definition: A disorder characterization | ed by occlusion of a vessel by a th | rombus that has migrated from a | distal site via the blood stream. | | 1 |
| Vasculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening; evidence of peripheral or visceral ischemia; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the w | all of a vessel. | | | |
| Visceral arterial ischemia | - | Brief (<24 hrs) episode of ischemia managed medically and without permanent deficit | Prolonged (>=24 hrs) or recurring symptoms and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characterize | ed by a decrease in blood supply | due to narrowing or blockage of a | visceral (mesenteric) artery. | | |
| Vascular disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |







NIH Publication No. 09-5410 Revised June 2010 Reprinted June 2010



## APPENDIX D. STANDARDIZED DEFINITIONS FOR CARDIOVASCULAR ENDPOINT EVENTS

| Event | Definitions |
|---|---|
| Cardiovascular (CV) Death: | |
| Death due to Acute MI | Death due to Acute MI refers to a death by any CV mechanism (eg, arrhythmia, sudden death, HF, stroke, pulmonary embolus, peripheral arterial disease) ≤30 days <sup>a</sup> after a MI related to the immediate consequences of the MI, such as progressive HF or recalcitrant arrhythmia. There may be assessable mechanisms of CV death during this time period, but for simplicity, if the CV death occurs ≤30 days of the MI, it will be considered a death due to MI. |
| | Acute MI should be verified to the extent possible by the diagnostic criteria outlined for acute MI (Clinical Data Interchange Standards Consortium [CDISC], Chapter 4) or by autopsy findings showing recent MI or recent coronary thrombosis. |
| | Death resulting from a procedure to treat a MI (percutaneous coronary intervention (PCI), coronary artery bypass graft surgery [CABG]), or to treat a complication resulting from MI, should also be considered death due to acute MI. |
| | Death resulting from an elective coronary procedure to treat myocardial ischemia (ie, chronic stable angina) or death due to a MI that occurs as a direct consequence of a CV investigation/procedure/operation should be considered as a death due to a CV procedure. |

| Event | Definitions |
|---|---|
| Sudden Cardiac Death | Sudden Cardiac Death refers to a death that occurs unexpectedly, not following an acute MI, and includes the following deaths: |
| | a. Death witnessed and occurring without new or worsening symptoms |
| | b. Death witnessed within 60 minutes of the onset of new or worsening cardiac symptoms, unless the symptoms suggest acute MI |
| | <ul> <li>Death witnessed and attributed to an identified arrhythmia (eg, captured on an electrocardiographic<br/>(ECG) recording, witnessed on a monitor, or unwitnessed but found on implantable cardioverter-<br/>defibrillator review)</li> </ul> |
| | <ul> <li>d. Death after unsuccessful resuscitation from cardiac arrest (eg, implantable cardioverter defibrillator<br/>(ICD) unresponsive sudden cardiac death, pulseless electrical activity arrest)</li> </ul> |
| | e. Death after successful resuscitation from cardiac arrest and without identification of a specific cardiac or non-cardiac etiology |
| | f. Unwitnessed death in a subject seen alive and clinically stable ≤24 hours prior to being found dead without any evidence supporting a specific non-CV cause of death (information regarding the subject's clinical status preceding death should be provided, if available). |
| | Unless additional information suggests an alternate specific cause of death (eg, death due to Other CV Causes), if a subject is seen alive ≤ 24 hours of being found dead, sudden cardiac death (criterion f above) should be recorded. For subjects who were not observed alive within 24 hours of death, undetermined cause of death should be recorded (eg, a subject found dead in bed, but who had not been seen by family for several days). |
| Death due to HF | Death due to HF refers to a death in association with clinically worsening symptoms and/or signs of HF regardless of HF etiology (CDISC, Chapter 7). Deaths due to HF can have various etiologies, including single or recurrent MIs, ischemic or non-ischemic cardiomyopathy, hypertension, or valvular disease. |
| Death due to Stroke | Death due to Stroke refers to death after a stroke (hemorrhagic, ischemic, or undetermined) that is either a direct consequence of the stroke or a complication of the stroke. Acute stroke should be verified to the extent possible by the diagnostic criteria outlined for stroke (CDISC, Chapter 6). |
| Death due to CV Procedures | Death due to CV Procedures refers to death caused by the immediate complications of a cardiac procedure. |
| Death due to CV Hemorrhage | Death due to CV Hemorrhage refers to death related to hemorrhage such as a non-stroke intracranial hemorrhage (CDISC, Chapter 6), non-procedural or non-traumatic vascular rupture (eg, aortic aneurysm), or hemorrhage causing cardiac tamponade. |
| Death due to Other CV Causes | Death due to Other CV Causes refers to a CV death not included in the above categories but with a specific, known cause (eg, pulmonary embolism or peripheral arterial disease). |

Version 4: 19 Dec 2016 Protocol 747-209


| Event | Definitions |
|---|---|
| Non-CV Death: | |
| The following is a suggested list of non-CV causes of death: | Non-CV death is defined as any death with a specific cause that is not thought to be CV in nature, as listed in CDISC Chapter 1, or as listed for CV Death. |
| <ul> <li>Pulmonary</li> </ul> | |
| • Renal | |
| <ul> <li>Gastrointestinal</li> </ul> | |
| <ul> <li>Hepatobiliary</li> </ul> | |
| <ul> <li>Pancreatic</li> </ul> | |
| <ul> <li>Infection (includes sepsis)</li> </ul> | |
| <ul> <li>Inflammatory (eg, Systemic<br/>Inflammatory Response<br/>Syndrome (SIRS) / immune<br/>(including autoimmune; may<br/>include anaphylaxis from<br/>environmental [eg, food]<br/>allergies)</li> </ul> | |
| <ul> <li>Hemorrhage that is neither CV<br/>bleeding nor a stroke (see<br/>Chapter 1, Section 6, and<br/>Chapter 6)</li> </ul> | |
| <ul> <li>Non-CV procedure or surgery</li> </ul> | |
| • Trauma | |
| • Suicide | |
| <ul> <li>Non-prescription drug reaction<br/>or overdose</li> </ul> | |
| <ul> <li>Prescription drug reaction or<br/>overdose (may include<br/>anaphylaxis)</li> </ul> | |
| <ul> <li>Neurological (non-CV)</li> </ul> | |
| <ul> <li>Malignancy</li> </ul> | |
| • Other non-CV | |

| Event | Definitions |
|---|---|
| <b>Undetermined Cause of Death:</b> | |
| Undetermined Cause of Death (will be classified as a CV death) | Undetermined cause of death refers to a death not attributable to one of the above categories of CV death or is due to a non-CV cause. Inability to classify the cause of death may be due to lack of information (eg, the only available information is "subject died") or there is insufficient supporting information or detail to assign the cause of death. In general, most deaths should be classifiable as CV or non-CV, and the use of this category of death, therefore, should be discouraged and should apply to few subjects in well-run clinical trials. |
| Cardiovascular Events: | |
| Myocardial Infarction <sup>b</sup> | a) <u>Clinical Presentation</u> |
| | The clinical presentation should be consistent with diagnosis of myocardial ischemia and infarction. Other findings that might support the diagnosis of MI should be taken into account because a number of conditions are associated with elevations in cardiac biomarkers (eg, trauma, surgery, pacing, ablation, HF, hypertrophic cardiomyopathy, pulmonary embolism, severe pulmonary hypertension, stroke or subarachnoid hemorrhage, infiltrative and inflammatory disorders of cardiac muscle, drug toxicity, burns, critical illness, extreme exertion, and chronic kidney disease). |
| | Supporting information can also be considered from myocardial imaging and coronary imaging. The totality of the data may help differentiate acute MI from the background disease process. |
| | b) <u>Biomarker Elevations</u> |
| | For cardiac biomarkers, laboratories should report an upper reference limit (URL). If the ninety-ninth percentile of the URL from the respective laboratory performing the assay is not available, then the URL for myocardial necrosis from the laboratory should be used. If the ninety-ninth percentile of the URL or the URL for myocardial necrosis is not available, the MI decision limit for the particular laboratory should be used as the URL. Laboratories can also report both the ninety-ninth percentile of the upper reference limit and the MI decision limit. Reference limits from the laboratory performing the assay are preferred over the manufacturer's listed reference limits in an assay's instructions for use. In general, troponins are preferred. Creatine kinase-myocardial band (CK-MB) should be used if troponins are not available, and total creatine kinase (CK) may be used in the absence of CK-MB and troponin. |
| | For MI subtypes, different biomarker elevations for CK, CK-MB, or troponin will be required. The specific criteria will be referenced to the URL. |
| | Since it is not practical to stipulate the use of a single biomarker or assay, the locally available results are to be used as the basis for adjudication. However, if possible, using the same cardiac biomarker assay and preferably, a core laboratory, for all measurements reduces inter-assay variability. |
| | Since the prognostic significance of different types of MIs (eg, periprocedural MI versus spontaneous MI) may be different, outcomes for these subsets of subjects may be evaluated separately. |

| Event | Definitions |
|---|---|
| | c) <u>ECG Changes</u> |
| | Electrocardiographic changes can be used to support or confirm a MI. Supporting evidence may be ischemic changes and confirmatory information may be new Q waves. |
| | ECG manifestations of acute myocardial ischemia (in absence of left ventricular hypertrophy [LVH] and left bundle branch block [LBBB]) include: |
| | • ST elevation: New ST elevation at the J point in two contiguous leads with the cut-points: ≥0.1 mV in all leads other than leads V2-V3 where the following cut-points apply: ≥0.2 mV in men ≥40 years (≥0.25 mV in men <40 years) or ≥0.15 mV in women |
| | <ul> <li>ST depression and T-wave changes: New horizontal or down-sloping ST depression ≥0.05 mV in two contiguous leads and/or new T inversion ≥ 0.1 mV in two contiguous leads with prominent R wave or R/S ratio &gt;1.</li> </ul> |
| | The above ECG criteria illustrate patterns consistent with myocardial ischemia. In subjects with abnormal biomarkers, it is recognized that lesser ECG abnormalities may represent an ischemic response and may be accepted under the category of abnormal ECG findings. |
| | Criteria for pathological Q-wave |
| | <ul> <li>Any Q-wave in leads V2-V3 ≥0.02 seconds or QS complex in leads V2 and V3</li> </ul> |
| | <ul> <li>Q-wave ≥0.03 seconds and ≥0.1 mV deep or QS complex in leads I, II, aVL, aVF, or V4-V6 in any two leads of a contiguous lead grouping (I, aVL; V1-V6; II, III, and aVF)<sup>c</sup></li> </ul> |
| | ECG changes associated with prior MI |
| | <ul> <li>Pathological Q-waves, as defined above</li> </ul> |
| | <ul> <li>R-wave ≥0.04 seconds in V1-V2 and R/S ≥1 with a concordant positive T-wave in the absence of a conduction defect</li> </ul> |
| | • Criteria for prior MI: Any one of the following criteria meets the diagnosis for prior MI: |
| | <ul> <li>Pathological Q waves with or without symptoms in the absence of non-ischemic causes</li> </ul> |
| | <ul> <li>Imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in<br/>the absence of a non-ischemic cause</li> </ul> |
| | Pathological findings of a prior myocardial infarction |
| Event | Definitions | | |
|---|---|--|--|
| Hospitalization for Unstable Angina | Unstable angina requiring hospitalization is defined as: 1. Ischemic discomfort (angina, or symptoms thought to be equivalent) ≥10 minutes in duration occurring | | |
| | <ul> <li>at rest, or</li> <li>in an accelerating pattern with frequent episodes associated with progressively decreased exercise capacity.</li> </ul> AND | | |
| | 2. Prompting an unscheduled hospitalization within 24 hours of the most recent symptoms. Hospitalization is defined as an admission to an inpatient unit or a visit to an emergency department that results in at least a 24 hour stay (or a change in calendar date if the hospital admission or discharge times are not available). | | |
| | <ul> <li>AND</li> <li>3. At least one of the following:</li> <li>a. New or worsening ST or T wave changes on resting ECG (in the absence of confounders, such as LBBB or LVH)</li> </ul> | | |
| | • Transient ST elevation (duration <20 minutes) New ST elevation at the J point in two contiguous leads with the cut-points: ≥0.1 mV in all leads other than leads V2-V3 where the following cut-points apply: ≥0.2 mV in men ≥40 years (≥0.25 mV in men <40 years) or ≥0.15 mV in women. | | |
| | <ul> <li>ST depression and T-wave changes</li> <li>New horizontal or down-sloping ST depression ≥0.05 mV in two contiguous leads and/or new T inversion ≥0.3 mV in two contiguous leads with prominent R wave or R/S ratio &gt;1.</li> </ul> | | |
| | <ul> <li>b. Definite evidence of inducible myocardial ischemia event as demonstrated by:</li> <li>• an early positive exercise stress test, defined as ST elevation or ≥2 mm ST depression prior to 5 mets OR</li> </ul> | | |
| | <ul> <li>stress echocardiography (reversible wall motion abnormality) OR</li> <li>myocardial scintigraphy (reversible perfusion defect), OR</li> </ul> | | |
| | <ul> <li>magnetic resonance imaging (MRI; myocardial perfusion deficit under pharmacologic stress).</li> <li>And believed to be responsible for the myocardial ischemic symptoms/signs.</li> <li>c. Angiographic evidence of new or worse ≥70% lesion (≥50% for left main lesion) and/or thrombus</li> </ul> | | |
| | in an epicardial coronary artery that is believed to be responsible for the myocardial ischemic symptoms/signs. | | |

| Event | Definitions | | |
|---|---|---|---|
| | d. Need for coronary revascularization procedure (PCI or CABG) for the presumed culprit lesion(s). This criterion would be fulfilled if revascularization was undertaken during the unscheduled hospitalization, or subsequent to transfer to another institution without interceding home discharge. AND | | |
| | Negative cardiac biomarkers and no evidence of acute MI | | |
| Transient Ischemic Attack (TIA) | | | as a transient episode of focal neurological dysfunction caused by brain, spinal cord, or retinal ut acute infarction. |
| <b>Stroke</b> (Includes Ischemic Stroke, Hemorrhagic Stroke, Undetermined | | | d as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or injury as a result of hemorrhage or infarction. |
| Stroke, or Stroke Disability) | <b>A. Ischemic Stroke:</b> Ischemic stroke is defined as an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of central nervous system tissue. | | |
| | | Hemorrhage may be a consequence of ischemic stroke. In this situation, the stroke is an ischemic stroke with hemorrhagic transformation and not a hemorrhagic stroke. | |
| | В. | <b>B. Hemorrhagic Stroke:</b> Hemorrhagic stroke is defined as an acute episode of focal or global cerebral or spinal dysfunction caused by intraparenchymal, intraventricular, or subarachnoid hemorrhage. | |
| | C. Undetermined Stroke: Undetermined stroke is defined as an acute episode of focal or global neurological dysfunction caused by presumed brain, spinal cord, or retinal vascular injury as a reshemorrhage or infarction but with insufficient information to allow categorization as A or B. | | |
| | | | ty: Disability should be measured by a reliable and valid scale in all cases, typically at each visit or the event. For example, the modified Rankin Scale may be used to address this requirement: |
| | | Scale | Disability |
| | | 0 | No symptoms at all |
| | | 1 | No significant disability despite symptoms; able to carry out all usual duties and activities |
| | | 2 | Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance |
| | | 3 | Moderate disability; requiring some help, but able to walk without assistance |
| | | 4 | Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance |
| | | 5 | Severe disability; bedridden, incontinent and requiring constant nursing care and attention |
| | | 6 | Dead |

| Event | Definitions |
|---|---|
| Heart Failure (A HF event includes | A HF hospitalization is defined as an event that meets ALL of the following criteria: |
| hospitalization for HF and may include urgent outpatient visits) | 1. The subject is admitted to the hospital with a primary diagnosis of HF |
| urgent outpatient visits) | 2. The subject's length-of-stay in hospital extends for at least 24 hours (or a change in calendar date if the hospital admission and discharge times are unavailable) |
| | 3. The subject exhibits documented new or worsening symptoms due to HF on presentation, including at least ONE of the following: |
| | Dyspnea (dyspnea with exertion, dyspnea at rest, orthopnea, paroxysmal nocturnal dyspnea) |
| | Decreased exercise tolerance |
| | Fatigue |
| | Other symptoms of worsened end-organ perfusion or volume overload (must be specified and described by the protocol) |
| | 4. The subject has objective evidence of new or worsening HF, consisting of at least TWO physical examination findings OR one physical examination finding and at least ONE laboratory criterion), including: |
| | a. Physical examination findings considered to be due to HF, including new or worsened: i.Peripheral edema |
| | ii.Increasing abdominal distention or ascites (in the absence of primary hepatic disease) iii.Pulmonary rales/crackles/crepitations |
| | iv.Increased jugular venous pressure and/or hepatojugular reflux |
| | v.S <sub>3</sub> gallop |
| | vi.Clinically significant or rapid weight gain thought to be related to fluid retention |
| | <ul> <li>Laboratory evidence of new or worsening HF, if obtained within 24 hours of presentation,<br/>including:</li> </ul> |
| | <ol> <li>Increased B-type natriuretic peptide (BNP)/ N-terminal pro-BNP (NT pro-BNP) concentrations consistent with decompensation of HF (such as BNP &gt; 500 pg/mL or NT- proBNP &gt;2,000 pg/mL). In subjects with chronically elevated natriuretic peptides, a significant increase should be noted above baseline.</li> </ol> |
| | ii.Radiological evidence of pulmonary congestion |

| Event | Definitions |
|---|---|
| | iii. Non-invasive diagnostic evidence of clinically significant elevated left- or right-sided ventricular filling pressure or low cardiac output. For example, ECG criteria could include: E/e' >15 or D-dominant pulmonary venous inflow pattern, plethoric inferior vena cava with minimal collapse on inspiration, or decreased left ventricular outflow tract (LVOT) minute stroke distance (time velocity integral [TVI]) |
| | OR |
| | iv. Invasive diagnostic evidence with right heart catheterization showing a pulmonary capillary wedge pressure (pulmonary artery occlusion pressure) ≥18 mmHg, central venous pressure ≥12 mmHg, or a cardiac index <2.2 L/min/m <sup>2</sup> |
| | Note: All results from diagnostic tests should be reported, if available, even if they do not meet the above criteria, because they provide important information for the adjudication of these events. |
| | 5. The subject receives initiation or intensification of treatment specifically for HF, including at least ONE of the following: |
| | a. Augmentation in oral diuretic therapy |
| | b. Intravenous diuretic or vasoactive agent (eg, inotrope, vasopressor, or vasodilator) |
| | c. Mechanical or surgical intervention, including: |
| | <ul> <li>Mechanical circulatory support (eg, intra-aortic balloon pump, ventricular assist device,<br/>extracorporeal membrane oxygenation, total artificial heart)</li> </ul> |
| | ii.Mechanical fluid removal (eg, ultrafiltration, hemofiltration, dialysis) |
| | An urgent HF visit is defined as an event that meets all of the following: |
| | 6. The subject has an urgent, unscheduled office/practice or emergency department visit for a primary diagnosis of HF, but not meeting the criteria for a HF hospitalization (i.e. urgent outpatient visit) |
| | 7. All signs and symptoms for HF hospitalization (ie, symptoms and physical examination findings/laboratory evidence of new or worsening HF, as indicated above) must be met |
| | 8. The subject receives initiation or intensification of treatment specifically for HF, as detailed in the above section with the exception of oral diuretic therapy, which will not be sufficient. |

| Event | Definitions |
|---|---|
| Interventional Cardiology: Clinical De | efinitions |
| Clinically-Driven Target Lesion<br>Revascularization: | Revascularization is clinically-driven if the target lesion diameter stenosis is >50% by quantitative coronary angiography (QCA) and the subject has clinical or functional ischemia which cannot be explained by another native coronary or bypass graft lesion. Clinical or functional ischemia includes any of the following: |
| | a. A history of angina pectoris, presumably related to the target vessel |
| | <ul> <li>Objective signs of ischemia at rest (electrocardiographic changes) or during exercise test (or<br/>equivalent), presumably related to the target vessel</li> </ul> |
| | c. Abnormal results of any invasive functional diagnostic test [e.g., coronary flow reserve (CFR) or fractional flow reserve (FFR)] |
| | <u>Comment</u> : Target lesion revascularization of a >70% diameter stenosis by QCA in the absence of the above signs or symptoms may be considered clinically-driven. |
| | <u>Comment</u> : In the absence of QCA data or if a $\leq$ 50% stenosis is present, TLR may be considered clinically-driven by the Adjudication Committee (AC) if severe ischemic signs and symptoms attributed to the target lesion are present. |
| Non-Target Lesion and Non-Target Lesion Revascularization: | A lesion for which revascularization is not attempted or one in which revascularization is performed using a non-study device, respectively. |
| Non-Target Vessel and Non-Target Vessel Revascularization: | A vessel for which revascularization is not attempted or one in which revascularization is performed using a non-study device, respectively. |
| Percutaneous Coronary Intervention (PCI) Status: | a. <b>Elective:</b> The procedure can be performed on an outpatient basis or during a subsequent hospitalization without significant risk of MI or death. For stable inpatients, the procedure is being performed during this hospitalization for convenience and ease of scheduling and <b>NOT</b> because the subject's clinical situation demands the procedure prior to discharge. |
| | b. <b>Urgent:</b> The procedure should be performed on an inpatient basis and prior to discharge because of significant concerns that there is risk of myocardial ischemia, MI, and/or death. Subjects who are outpatients or in the emergency department at the time that the cardiac catheterization is requested would warrant hospital admission based on their clinical presentation. |
| | c. <b>Emergency:</b> The procedure should be performed as soon as possible because of substantial concerns that ongoing myocardial ischemia and/or MI could lead to death. "As soon as possible" refers to a subject whis of sufficient acuity that one would cancel a scheduled case to perform this procedure immediately in the next available room during business hours, or one would activate the on-call team were this to occur during off-hours. |

| Event | Definitions |
|---|---|
| | d. <b>Salvage:</b> The procedure is a last resort. The subject is in cardiogenic shock when the PCI begins (ie, the time at which the first guide wire or intracoronary device is introduced into a coronary artery or bypass graft for the purpose of mechanical revascularization) <b>OR</b> within the last ten minutes prior to the start of the case or during the diagnostic portion of the case, the subject has also received chest compressions or has been on unanticipated circulatory support (eg, intra-aortic balloon pump, extracorporeal membrane oxygenation, or cardiopulmonary support). |
| Percutaneous Coronary Intervention (PCI): | Placement of an angioplasty guide wire, balloon, or other device (e.g., stent, atherectomy catheter, brachytherapy delivery device, or thrombectomy catheter) into a native coronary artery or coronary artery bypass graft for the purpose of mechanical coronary revascularization. In the assessment of the severity of coronary lesions with the use of intravascular ultrasound, coronary flow reserve (CFR), or fractional flow reserve (FFR), insertion of a guide wire will <b>NOT</b> be considered PCI. |
| Procedural Success: | Achievement of <30 % residual diameter stenosis of the target lesion assessed by visual inspection or QCA and no in-hospital major adverse cardiac events (MACE, a composite of death, MI, or repeat coronary revascularization of the target lesion). Ideally, the assessment of the residual stenosis at the end of the procedure should be performed by an angiographic core laboratory. |
| | <b>Comment:</b> For some device interventions (eg, balloon angioplasty), achievement of <50% diameter stenosis by visual inspection or QCA is an acceptable definition for procedural success. |
| Target Lesion: | Any lesion treated or attempted to be treated during the PCI with the study device. The target lesion includes the arterial segment treated with the study device (stent, in most cases) plus 5 mm proximal and 5 mm distal to the treatment site. |
| Target Lesion Failure (TLF): | The composite of ischemia-driven revascularization of the target lesion, MI related to the target vessel, or cardiac death related to the target vessel. If it cannot be determined with certainty whether the MI or death was related to the target vessel, it is considered a TLF. |
| Target Lesion Revascularization (TLR): | Any repeat percutaneous intervention of the target lesion (including 5 mm proximal and 5 mm distal to the target lesion) or surgical bypass of the target vessel performed for restenosis or other complication involving the target lesion. In the assessment of TLR, angiograms should be assessed by an angiographic core laborator (if designated) and made available to the AC for review upon request. |
| Target Vessel: | A major native coronary artery (eg, left main coronary artery, left anterior descending coronary artery, left circumflex coronary artery, or right coronary artery) or bypass graft containing the target lesion. A native coronary artery target vessel includes the arterial segments upstream and downstream to the target lesion plus major side branches. |
| Target Vessel Failure (TVF): | The composite of ischemia-driven revascularization of the target vessel, MI related to the target vessel, or cardiac death related to the target vessel. If it cannot be determined with certainty whether the MI or death was related to the target vessel, it is considered a TVF. |

| Event | Definitions | |
|---|---|---|
| Target Vessel, Non-Target Lesion, and Target Vessel, Non-Target Lesion Revascularization: | Any lesion or revascularization of a lesion in the target vessel other than the target lesion, respectively. | |
| Target Vessel Revascularization (TVR): | Any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. In the assessment of TVR, angiograms should be assessed by an angiographic core laboratory (if designated) and made available to the CEC for review upon request. | |
| Vascular Complications: | Access site hematoma: Development of a new, localized collection of blood at a vascular access site sufficient to produce a palpable mass within 72 hours of a procedure. | |
| | | ala: Development of a new, unintended communication between an artery and a vascular access site within 72 hours of a procedure. |
| | • <b>Peripheral ischemia:</b> Development of new arterial insufficiency sufficient to produce clinical signs or symptoms of ischemia (pallor, pain, paresthesia) distal to a vascular access site within 72 hours of a procedure. | |
| | • <b>Peripheral nerve injury:</b> Development of new sensory or motor loss of peripheral nerve function from external nerve compression (e.g., as a result of positioning during a procedure), or internal compression or direct nerve damage from the procedure, occurring within 72 hours of a procedure. | |
| | • <b>Pseudoaneurysm:</b> Development of a new localized collection of blood with a persistent communication (neck) originating at a vascular access site and occurring within 72h of a procedure. | |
| | • <b>Retroperitoneal hemorrhage:</b> Development of new bleeding into the retroperitoneal space originating at a vascular access site and occurring within 72 hours of a procedure. | |
| Interventional Cardiology: Angiograp | ohic Definitions | |
| Abrupt Closure: | New intra-procedural severely reduced flow (TIMI grade 0-1) within the target vessel that persists and requires intervention by stenting or other treatment, or results in MI or death. Abrupt closure requires an association with a vascular dissection, thrombus, or severe spasm at the treatment site or within the instrumented vessel. | |
| <b>Coronary Lesions Treated</b> | Coronary Artery<br>Segments | Definitions |
| | Right coronary artery ostium | Origin of the right coronary artery, including the first 3 mm of the artery |
| | Proximal right coronary artery | Proximal portion of the right coronary artery, from the ostium of the right coronary artery to the origin of the first right ventricular branch (pRCA) |

| Event | | Definitions |
|---|---|---|
| | Mid right coronary artery | Middle portion of the right coronary artery, from the origin of the first right ventricular branch to the acute margin (mRCA) |
| | Distal right coronary artery | Distal portion of the right coronary artery, from the acute margin to the origin of the posterior descending artery (dRCA) |
| | Right posterior descending artery | In right dominant and mixed circulations, the vessel that runs in the posterior interventricular groove and supplies septal perforator branches (PDA) |
| | Posterolateral segmental artery | In right dominant circulations, the distal continuation of the right coronary artery in the posterior atrioventricular groove after the origin of the right posterior descending artery (PLSA) |
| | First right posterolateral branch | In right dominant circulations, the first posterolateral branch originating from the right posterior atrioventricular artery (RPL1) |
| | Second right posterolateral branch | In right dominant circulations, the second posterolateral branch originating from the right posterior atrioventricular artery (RPL2) |
| | Third right posterolateral branch | In right dominant circulations, the third posterolateral branch originating from the right posterior atrioventricular artery (RPL3) |
| | Posterior descending septal perforator | Septal perforator vessel originating from the posterior descending artery |
| | Right ventricular branch | Branch arising from the right coronary artery to supply the right ventricular wall (RV) |
| | Left main coronary artery ostium | Origin of the left coronary artery, including the first 3 mm of the artery |
| | Left main coronary artery body | Body of the left main coronary artery, from the ostium to the bifurcation (LM) |
| | Left main coronary artery bifucation | Distal end of the left main, including the terminal 3 mm through the bifurcation of the left main into the left anterior descending and left circumflex arteries |
| | Left anterior descending artery ostium | Origin of the left anterior descending coronary artery, including the first 3 mm of the artery |
| | Proximal left anterior descending artery | Proximal portion of the left anterior descending coronary artery, from the ostium to the origin of the first septal (pLAD) |
| | Mid left anterior descending artery | Middle portion of the left anterior descending coronary artery, from the origin of the first septal artery to the origin of the third septal artery (mLAD) |

| Event | Definitions | |
|---|---|---|
| | Distal left anterior descending artery | Distal portion of the left anterior descending coronary artery, from the origin of the third septal artery to the terminus (dLAD) |
| | First diagonal branch | First of the three longest branches originating from the left anterior descending artery to supply the anterolateral wall of the left ventricle (D1) |
| | First diagonal lateral branch | Branch of the first diagonal branch |
| | Second diagonal branch | Second of the three longest branches originating from the left anterior descending artery to supply the anterolateral wall of the left ventricle (D2) |
| | Second diagonal lateral branch | Branch of the second diagonal branch |
| | Third diagonal branch | Third of the three longest branches originating from the left anterior descending artery to supply the anterolateral wall of the left ventricle (D3) |
| | Third diagonal lateral branch | Branch of the third diagonal branch |
| | Anterior descending septal perforator | Septal perforator vessel originating from the left anterior descending artery to supply the interventricular septum |
| | Left circumflex artery ostium | Origin of the left circumflex coronary artery, including the first 3 mm of the artery |
| | Proximal left circumflex artery | Proximal portion of the left circumflex coronary artery, from the ostium to the origin (or the nominal location of) the first marginal branch (pLCX) |
| | Mid left circumflex artery | Middle portion of the left circumflex coronary artery, from the origins of (or nominal locations of) the first marginal to the second marginal (mLCX) |
| | Distal left circumflex artery | Distal portion of the left circumflex coronary artery, from the origin of (or the nominal location of) the second marginal to the terminus (in right dominant systems), or to the origin of the 1st left posterolateral in all other dominance systems (dLCX) |
| | First obtuse marginal branch | First of the three longest branches originating from the left circumflex artery to supply the lateral wall of the left ventricle (OM1) |
| | First obtuse marginal lateral branch | Branch of the first marginal branch |
| | Second obtuse marginal branch | Second of the three longest branches originating from the left circumflex artery to supply the lateral wall of the left ventricle (OM2) |

| Event | Definitions | |
|---|---|---|
| | Second obtuse marginal lateral branch | Branch of the second marginal branch |
| | Third obtuse marginal branch | Third of the three longest branches originating from the left circumflex artery to supply the lateral wall of the left ventricle (OM3) |
| | Third obtuse marginal lateral branch | Branch of the third marginal branch |
| | Left atrioventricular artery | In left dominant and mixed circulations, the distal continuation of the left circumflex coronary artery in the posterior atrioventricular groove |
| | Left posterior descending artery | In left dominant circulations, the vessel that arises from the distal continuation of the left atrioventricular artery, travels in the posterior interventricular groove, and supplies septal perforator branches (LPDA) |
| | First left posterolateral branch | In left dominant and mixed circulations, the first posterolateral branch originating from the posterior atrioventricular left circumflex artery (LPL1) |
| | Second left posterolateral branch | In left dominant and mixed circulations, the second posterolateral branch originating from the posterior atrioventricular left circumflex artery (LPL2) |
| | Third left posterolateral branch | In left dominant and mixed circulations, the third posterolateral branch originating from the posterior atrioventricular left circumflex artery (LPL3) |
| | Ramus intermedius branch | Branch vessel whose origin bisects the origins of the left anterior descending and circumflex arteries (RI) |
| | Ramus intermedius lateral branch | Branch of the ramus intermedius branch |
| Dissection: | Based on the National Hea | rt, Lung, and Blood Institute (NHLBI) Dissection Classification System: |
| | Grade A: Minor radio clearance | lucencies within the lumen during contrast injection with no persistence after dye |
| | Grade B: Parallel trac<br>persistence after dye cl | ts or double lumen separated by a radiolucent area during contrast injection with no earance |
| | Grade C: Extralumina | ll cap with persistence of contrast after dye clearance from the lumen |
| | Grade D: Spiral lumin | nal filling defect with delayed but complete distal flow |
| | • Grade E: New persiste | ent filling defect with delayed antegrade flow |
| | | oes with total coronary occlusion and no distal antegrade flow ions may represent thrombus |

| Event | Definitions |
|---|---|
| Late Loss: | Minimum lumen diameter (MLD) assessed at follow-up angiography minus the MLD assessed immediately after the index procedure. MLDs are measured by QCA. |
| Minimum Lumen Diameter (MLD): | The mean minimum lumen diameter (typically measured in-lesion, in-stent, and in-segment) derived from two orthogonal views by QCA. |
| No Reflow: | An acute reduction in coronary flow (TIMI grade 0-1) in the absence of dissection, thrombus, spasm, or high-grade residual stenosis at the original target lesion. |
| Percent Diameter Stenosis (% DS): | The value calculated as 100 x (1 – MLD/RVD) using the mean values determined by QCA from two orthogonal views (when possible). |
| Reference Vessel Diameter (RVD): | Defined as the average of normal segments within 10 mm proximal and 10 mm distal to the target lesion from two orthogonal views using QCA. |
| Restenosis: | Re-narrowing of the vessel following the treatment of a prior stenosis |
| | • <b>Binary restenosis:</b> A diameter stenosis of > 50% at the previously treated lesion site, including the originally treated site plus the adjacent vascular segments 5 mm proximal and 5 mm distal to the site. |
| | • In-stent restenosis (ISR): A previously stented lesion with a > 50% diameter stenosis. |
| Thrombus (Angiographic): | A discrete, mobile, intraluminal filling defect with defined borders with or without associated contrast staining. |
| TIMI (Thrombolysis in Myocardial | • Grade 0 (no perfusion): There is no antegrade flow beyond the point of occlusion. |
| Infarction) Flow Grades: | <ul> <li>Grade 1 (penetration without perfusion): The contrast material passes beyond the area of obstruction but "hangs up" and fails to opacify the entire coronary bed distal to the obstruction for the duration of the cineangiographic filming sequence.</li> </ul> |
| | • Grade 2 (partial perfusion): The contrast material passes across the obstruction and opacifies the coronary bed distal to the obstruction. However, the rate of entry of contrast material into the vessel distal to the obstruction or its rate of clearance from the distal bed (or both) is perceptibly slower than its entry into or clearance from comparable areas not perfused by the previously occluded vessel (eg, the opposite coronary artery or the coronary bed proximal to the obstruction). |
| | • Grade 3 (complete perfusion): Antegrade flow into the bed distal to the obstruction occurs as promptly as antegrade flow into the bed proximal to the obstruction and clearance of contrast material from the involved bed is as rapid as from an uninvolved bed in the same vessel or the opposite artery. |
| Vessels | Left main coronary artery (LMCA) |
| | Left anterior descending artery (LAD) with septal and diagonal branches |

| Event | Definitions |
|---|---|
| | Left circumflex artery (LCX) with obtuse marginal branches |
| | Ramus intermedius artery |
| | • Right coronary artery (RCA) and any of its branches |
| | Posterior descending artery |
| | • Saphenous vein bypass graft(s) |
| | • Arterial bypass graft(s): Right internal mammary graft, left internal mammary graft, radial artery graft, and gastroepiploic artery graft. |
| Peripheral Vascular Intervention | |
| Peripheral Vascular Intervention (PVI): | Peripheral vascular intervention <sup>d</sup> is a catheter based or open surgical procedure designed to improve arterial or venous blood flow or otherwise modify or revise vascular conduits. Procedures may include, but are not limited to, percutaneous transluminal balloon angioplasty, stent placement, thrombectomy, embolectomy, atherectomy, dissection repair, aneurysm exclusion, treatment of dialysis conduits, placement of various devices, intravascular thrombolysis or other pharmacotherapies, and open surgical bypass or revision. |
| | In general, the intention to perform <i>percutaneous</i> peripheral vascular intervention is denoted by the insertion a guide wire into a peripheral artery or vein. |
| | The target vessel(s) and the type of revascularization procedure (e.g., surgical bypass, thrombectomy, endarterectomy, percutaneous transluminal angioplasty, stent placement, thromboembolectomy, and thrombolysis) should be specified and recorded. For the sake of simplicity, this definition applies to the extracranial carotid artery and other non-cardiac arteries and veins and excludes the intracranial vessels and lymphatics. |
| Procedural Success: | In the case of percutaneous intervention for obstructive lesions, procedural success is defined as the achievement of a satisfactory final residual diameter stenosis by angiography at the end of the procedure (and without flow limiting dissection or hemodynamically significant translesional pressure gradient). The specific parameter for final percent residual stenosis is typically between <30% and <50%; selection of the appropriate percentage may vary depending upon the specific intervention applied, the vascular territory, and anticipated or desired therapeutic response. Procedural success also implies absence of in-hospital major adverse events (eg, death, stroke, myocardial infarction, acute onset of limb ischemia, need for urgent/emergent vascular surgery, and other procedure-specific major adverse events). The balloon inflation, stent placement, or other therapeutic intervention may be preceded by use of adjunctive devices (eg, percutaneous mechanical thrombectomy, directional or rotational atherectomy, laser, and chronic total occlusion crossing device), as predefined in the protocol. |

| Event | Definitions |
|---|---|
| Procedural Status: Non-Elective and Elective: | e. <b>Non-Elective:</b> Non-elective procedures include emergent and urgent procedures. A non elective procedure is a procedure that is performed without delay, because there is clinical consensus that the procedure should occur imminently. Non-elective procedures imply a degree of instability of the subject, urgency of the medical condition, or instability of the threatening lesion. |
| | <ul> <li>Emergent: A procedure that is performed immediately because of the acute nature of the medical condition (e.g., acute limb ischemia, acute aortic dissection), and the increased morbidity or mortality associated with a temporal delay in treatment.</li> </ul> |
| | <ul> <li>Urgent: An urgent procedure is one that is not an emergency but is required to be performed on a timely basis (≤24 hrs) (e.g., a subject who has been stabilized following initial treatment of acute limb ischemia, and there is clinical consensus that a definitive procedure should occur within the next 24 hours).</li> </ul> |
| | f. <b>Elective:</b> An elective procedure is one that is scheduled and is performed on a subject with stable disease, or in whom there is no urgency and/or increased morbidity or mortality associated with a planned procedure. |
| Target Lesion: | A target lesion is any vascular segment treated or attempted to be treated during the trial procedure with the index device. The target lesion is the treated segment starting 10 mm proximal and ending 10 mm distal to the index device or therapy (stent, balloon, atherectomy catheter, or aortic stent-graft). |
| Target Vessel: | A target vessel is any vessel (eg, non-cardiac or non-intracranial) that contains the target lesion treated with the study device. The target vessel includes the target lesion as well as the entire length of native vessel upstream and downstream from the target lesion, including side branches. For the arteries of the leg, the vasculature is divided into 3 vessel "levels:" aorto-iliac, femoral-popliteal, and tibial-crural. |
| Non-Target Lesion and Non-Target<br>Lesion Revascularization: | A lesion for which revascularization is not attempted or one in which revascularization is performed using a non-study device, respectively. |
| Non-Target Vessel and Non-Target<br>Vessel Revascularization: | A vessel for which revascularization is not attempted or one in which revascularization is performed using a non-study device, respectively. |
| Target Vessel, Non-Target Lesion<br>and Target Vessel, Non-Target<br>Lesion Revascularization: | Any lesion or revascularization of a lesion in the target vessel other than the target lesion, respectively. |
| Target Lesion Revascularization (TLR): | Target lesion revascularization is any repeat intervention of the target lesion (including 10 mm proximal and 10 mm distal to the index device, as target lesion is defined above) or surgical intervention/bypass of the target vessel performed for restenosis or other complication involving the target lesion. In the assessment of TLR, angiograms should be assessed by an angiographic core laboratory (if designated). Angiograms (and core laboratory assessment thereof) and other source documentation should be made available to the CEC for review upon request. |

| Event | Definitions |
|---|---|
| Target Vessel Revascularization (TVR): | Target vessel revascularization is any repeat intervention or surgical bypass of any segment of the target vessel. In the assessment of TVR, angiograms should be assessed by an angiographic core laboratory (if designated). Angiograms (and core laboratory assessment thereof) and other source documentation should be made available to the CEC for review upon request. |
| Clinically-Driven Target Lesion<br>Revascularization: | Clinically-driven target lesion revascularization is defined as target lesion revascularization performed due to target lesion diameter stenosis >50% <b>AND</b> either evidence of clinical or functional ischemia (eg, recurrent/progressive intermittent claudication, critical limb ischemia) <b>OR</b> recurrence of the clinical syndrome for which the initial procedure was performed. Clinically-driven target lesion revascularization occurs in the absence of protocol-directed surveillance ultrasound or angiography. |
| Vessel Patency: | Vessel patency at a given time point will be determined by the absence of clinically-driven target lesion revascularization and/or absence of recurrent target lesion diameter stenosis >50% by imaging (eg, invasive angiography or most commonly, duplex ultrasonography). If patency data are incorporated within the primary endpoint of a clinical trial, the angiographic images or duplex ultrasonographic images should be assessed by appropriate core laboratories and made available to the AC for review upon request. |
| Restenosis: | Re-narrowing of the artery following the treatment of a prior stenosis |
| | • <b>Binary restenosis:</b> A diameter stenosis of >50% at the previously treated lesion site, including the originally treated site plus the adjacent vascular segments 10 mm proximal and 10 mm distal to the site (or as otherwise defined by the protocol, as noted above). |
| | • In-stent restenosis (ISR): A previously stented lesion that has >50% diameter stenosis. |

| Event | | Definitions |
|---|---|---|
| Stent Thrombosis | | |
| Stent Thrombosis: Timing | Stent thrombosis should be reported as a cumulative value over time and at the various individual time points as specified below. Time 0 is defined as the time point after the guiding catheter has been removed and the subject has left the cardiac catheterization laboratory. Stent Thrombosis: Timing | |
| | Acute stent thrombosis <sup>1</sup> | 0-24 hours post stent implantation |
| | Subacute stent thrombosis <sup>1</sup> | >24 hours – 30 days post stent implantation |
| | Late stent thrombosis <sup>2</sup> | >30 days – 1 year post stent implantation |
| | Very late stent thrombosis <sup>2</sup> | >1 year post stent implantation |
| | Acute or subacute can also be replaced by the term early stent thrombosis. Early stent thrombosis (0-30 days) will be used herein. Includes "primary" as well as "secondary" late stent thrombosis; "secondary" late stent thrombosis is a stent thrombosis after a target lesion revascularization. | |
| Stent Thrombosis Categories | <ol> <li>Definite Stent Thrombosis Definite stent thrombosis is considered to have occurred by either angiographic or pathological confirmation: a. Angiographic confirmation of stent thrombosis<sup>c</sup> </li> </ol> | |
| | <ul> <li>Angiographic confirmation of stent thrombosis<sup>c</sup></li> <li>The presence of a thrombus<sup>f</sup> that originates in the stent or in the segment 5 mm proximal or distal to the stent and presence of at least 1 of the following criteria within a 48-hour time window: <ul> <li>Acute onset of ischemic symptoms at rest</li> <li>New ischemic ECG changes that suggest acute ischemia</li> <li>Typical rise and fall in cardiac biomarkers (refer to definition of spontaneous MI)</li> <li>Nonocclusive thrombus: Intracoronary thrombus is defined as a (spheric, ovoid, or irregular) noncalcified filling defect or lucency surrounded by contrast material (on 3 sides or within a coronary stenosis) seen in multiple projections, or persistence of contrast material within the lumen, or a visible embolization of intraluminal material downstream</li> </ul> </li> </ul> | |
| | | ombus: TIMI 0 or TIMI 1 intrastent or proximal to a stent up to the most imal side branch or main branch (if originates from the side branch). |


| Event | Definitions |
|---|---|
| | <b>b.</b> Pathological Confirmation of Stent Thrombosis: Evidence of recent thrombus within the stent determined at autopsy or via examination of tissue retrieved following thrombectomy. |
| | 2. <b>Probable Stent Thrombosis:</b> Clinical definition of probable stent thrombosis is considered to have occurred after intracoronary stenting in the following cases: |
| | a. Any unexplained death within the first 30 days <sup>g</sup> |
| | b. Irrespective of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause |
| | <ol> <li>Possible Stent Thrombosis: Clinical definition of possible stent thrombosis is considered to have<br/>occurred with any unexplained death from 30 days after intracoronary stenting until end of trial<br/>follow-up.</li> </ol> |

<sup>&</sup>lt;sup>a</sup> The 30-day cut-off is arbitrary.

g For studies with ST-elevation MI population, one may consider the exclusion of unexplained death within 30 days as evidence of probable stent thrombosis.

Source: "Standardized Definitions for Cardiovascular and Stroke Endpoint Events in Clinical Trials," dated August 20, 2014, and available at the CDISC website (http://www.cdisc.org/system/files/all/standard/Draft%20Definitions%20for%20CDISC%20August%2020,%202014.pdf).

Note: CEC = Cardiovascular Events Committee, which is referred to in the body of the protocol as the CAC = Cardiovascular Adjudication Committee

<sup>&</sup>lt;sup>b</sup> 2012 Third Universal Definition of Myocardial Infarction.

<sup>&</sup>lt;sup>c</sup> The same criteria are used for supplemental leads V7-V9, and for the Cabrera frontal plane lead grouping.

<sup>&</sup>lt;sup>d</sup> Peripheral vascular disease includes veins, arteries, and lymphatics. However, for simplicity, this definition focuses on peripheral artery and venous interventions.

<sup>&</sup>lt;sup>e</sup> The incidental angiographic documentation of stent occlusion in the absence of clinical signs or symptoms is not considered a confirmed stent thrombosis (silent occlusion).

f Intracoronary thrombus.

| Event | Mechanism/Classification | Definitions |
|---|---|---|
| Event Hospitalization for Unstable Angina | <ol> <li>General Considerations</li> <li>Escalation of pharmacotherapy for ischemia, such as intravenous nitrates or increasing dosages of β-blockers, should be considered supportive but not diagnostic of unstable angina. However, a typical presentation and admission to the hospital with escalation of pharmacotherapy, without any of the additional findings listed under item 3 above, would be insufficient to support classification as hospitalization for unstable angina.</li> <li>If subjects are admitted with suspected unstable angina, and subsequent testing reveals a non-cardiac or non-ischemic etiology, this event should not be recorded as hospitalization for unstable</li> </ol> | <ul> <li>Unstable angina requiring hospitalization is defined as: <ol> <li>Ischemic discomfort (angina, or symptoms thought to be equivalent) ≥10 minutes in duration occurring</li> <li>at rest, or</li> <li>in an accelerating pattern with frequent episodes associated with progressively decreased exercise capacity.</li> </ol> </li> <li>AND</li> <li>Prompting an unscheduled hospitalization within 24 hours of the most recent symptoms. Hospitalization is defined as an admission to an inpatient unit or a visit to an emergency department that results in at least</li> </ul> |
| | angina. Potential ischemic events meeting the criteria for MI should not be adjudicated as unstable angina. 3. Planned hospitalization or rehospitalization for performance of an elective revascularization in subjects who do not fulfill the criteria for unstable angina should not be considered a hospitalization for unstable angina. • Hospitalization of a subject with stable exertional angina for coronary angiography and PCI that is prompted by a positive outpatient stress test should not be considered hospitalization for unstable angina. • Rehospitalization of a subject meeting the criteria for unstable angina who was stabilized, discharged, and subsequently readmitted for revascularization, | a 24 hour stay (or a change in calendar date if the hospital admission or discharge times are not available). AND 3. At least one of the following: a. New or worsening ST or T wave changes on resting ECG (in the absence of confounders, such as LBBB or LVH) • Transient ST elevation (duration <20 minutes) New ST elevation at the J point in two contiguous leads with the cutpoints: ≥0.1 mV in all leads other than leads V2-V3 where the following cut-points apply: ≥0.2 mV in men ≥40 years (≥0.25mV in men <40 years) or ≥0.15 mV in women. |


| Event | Mechanism/Classification | Definitions |
|---|---|---|
| Hospitalization for Unstable | does not constitute a second hospitalization for | ST depression and T-wave changes |
| Angina<br>(Continued) | unstable angina. A subject who undergoes an elective catheterization where incidental coronary artery disease is found and who subsequently undergoes coronary revascularization will not be considered as meeting the hospitalization for unstable angina endpoint. | • New horizontal or down-sloping ST depression ≥0.05 mV in two contiguous leads and/or new T inversion ≥0.3 mV in two contiguous leads with prominent R wave or R/S ratio >1. |
| | | <ul> <li>Definite evidence of inducible myocardial ischemia event as demonstrated by:</li> </ul> |
| | | • an early positive exercise stress test, defined as ST elevation or ≥2 mm ST depression prior to 5 mets OR |
| | | <ul> <li>stress echocardiography (reversible wall motion abnormality) OR</li> </ul> |
| | | <ul> <li>myocardial scintigraphy (reversible perfusion defect), OR</li> </ul> |
| | | <ul> <li>magnetic resonance imaging (MRI;<br/>myocardial perfusion deficit under<br/>pharmacologic stress).</li> </ul> |
| | | <ul> <li>And believed to be responsible for the<br/>myocardial ischemic symptoms/signs.</li> </ul> |
| | | <ul> <li>c. Angiographic evidence of new or worse ≥70% lesion (≥50% for left main lesion) and/or thrombus in an epicardial coronary artery that is believed to be responsible for the myocardial ischemic symptoms/signs.</li> </ul> |
| | | d. Need for coronary revascularization procedure (PCI or CABG) for the presumed culprit lesion(s). This criterion would be fulfilled if revascularization was undertaken during the unscheduled hospitalization, or subsequent to transfer to another institution without interceding home discharge. |

| Event | Mechanism/Classification | Definitions |
|---|---|---|
| | | AND AND Negative cardiac biomarkers and no evidence of acute MI |
| Transient Ischemic Attack (TIA) and Stroke | TIA | TIA is defined as a transient episode of focal neurological dysfunction caused by brain, spinal cord, or retinal ischemia, without acute infarction. |
| and stroke | Stroke Classification: | Stroke is defined as an acute episode of focal or global |
| | A. Ischemic Stroke | neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction. |
| | Ischemic stroke is defined as an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of central nervous system tissue. | |
| | Hemorrhage may be a consequence of ischemic stroke. In this situation, the stroke is an ischemic stroke with hemorrhagic transformation and not a hemorrhagic stroke. | |
| | B. Hemorrhagic Stroke | |
| | Hemorrhagic stroke is defined as an acute episode of focal or global cerebral or spinal dysfunction caused by intraparenchymal, intraventricular, or subarachnoid hemorrhage. | |
| | C. Undetermined Stroke | |
| | Undetermined stroke is defined as an acute episode of focal or global neurological dysfunction caused by presumed brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction but with insufficient information to allow categorization as A or B. | |


| Event | Mecha | anism/Classification | Definitions |
|---|---|---|---|
| Transient<br>Ischemic<br>Attack (TIA)<br>and Stroke<br>(Continued) | D. Stroke Disability Disability should be measured by a reliable and valid scale in all cases, typically at each visit and 90 days after the event. For example, the modified Rankin Scale may be used to address this requirement: | | · |
| | Scale | Disability | |
| | 0 | No symptoms at all | |
| | 1 | No significant disability despite symptoms; able to carry out all usual duties and activities | |
| | 2 | Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance | |
| | 3 | Moderate disability; requiring some help, but able to walk without assistance | |
| | 4 | Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance | |
| | 5 | Severe disability; bedridden, incontinent and requiring constant nursing care and attention | |
| | 6 | Dead | |


| Event | Mechanism/Classification | Definitions |
|---|---|---|
| HF Event : A HF event | | A HF hospitalization is defined as an event that meets ALL of the following criteria: |
| includes hospitalization for HF and may | | 1. The subject is admitted to the hospital with a primary diagnosis of HF |
| include urgent<br>outpatient<br>visits. HF<br>hospitalizations<br>should remain | | 2. The subject's length-of-stay in hospital extends for at least 24 hours (or a change in calendar date if the hospital admission and discharge times are unavailable) |
| delineated from<br>urgent visits. If<br>urgent visits are<br>included in the<br>HF endpoint, | | 3. The subject exhibits documented new or worsening symptoms due to HF on presentation, including at least ONE of the following: |
| the number of<br>urgent visits<br>needs to be<br>explicitly | | <ul> <li>Dyspnea (dyspnea with exertion, dyspnea at<br/>rest, orthopnea, paroxysmal nocturnal<br/>dyspnea)</li> </ul> |
| presented separately from | | Decreased exercise tolerance |
| the | | • Fatigue |
| hospitalizations. | | <ul> <li>Other symptoms of worsened end-organ<br/>perfusion or volume overload (must be<br/>specified and described by the protocol)</li> </ul> |
| | | 4. The subject has objective evidence of new or worsening HF, consisting of at least TWO physical examination findings OR one physical examination finding and at least ONE laboratory criterion), including: |
| | | a. Physical examination findings considered to be due to HF, including new or worsened: |
| | | i.Peripheral edema |


Version 4: 19 Dec 2016

| Event | Mechanism/Classification | Definitions |
|---|---|---|
| HF Event (Continued): | | ii.Increasing abdominal distention or ascites (in the absence of primary hepatic disease) |
| A HF event | | iii.Pulmonary rales/crackles/crepitations |
| includes<br>hospitalization<br>for HF and may | | iv.Increased jugular venous pressure and/or hepatojugular reflux |
| include urgent | | v.S <sub>3</sub> gallop |
| outpatient<br>visits. HF<br>hospitalizations | | vi.Clinically significant or rapid weight gain thought to be related to fluid retention |
| should remain<br>delineated from<br>urgent visits. If | | b. Laboratory evidence of new or worsening HF, if obtained within 24 hours of presentation, including: |
| urgent visits are included in the HF endpoint, the number of urgent visits needs to be explicitly presented | | i.Increased B-type natriuretic peptide (BNP)/ N-terminal pro-BNP (NT pro-BNP) concentrations consistent with decompensation of HF (such as BNP >500 pg/mL or NT-proBNP >2,000 pg/mL). In subjects with chronically elevated natriuretic peptides, a significant increase should be noted above baseline. |
| separately from the | | ii.Radiological evidence of pulmonary congestion |
| hospitalizations. | | iii.Non-invasive diagnostic evidence of clinically significant elevated left- or right-sided ventricular filling pressure or low cardiac output. For example, ECG criteria could include: E/e' >15 or D-dominant pulmonary venous inflow pattern, plethoric inferior vena cava with minimal collapse on inspiration, or decreased left ventricular outflow tract (LVOT) minute stroke distance (time velocity integral [TVI]) |
| | | OR |
| | | iv.Invasive diagnostic evidence with right heart catheterization showing a pulmonary capillary wedge pressure (pulmonary artery occlusion |

Protocol 747-209 Version 4: 19 Dec 2016


| Event | Mechanism/Classification | Definitions |
|---|---|---|
| HF Event (Continued): | | pressure) ≥18 mmHg, central venous pressure<br>≥12 mmHg, or a cardiac index <2.2 L/min/m <sup>2</sup> |
| A HF event includes hospitalization for HF and may | | Note: All results from diagnostic tests should be reported, if available, even if they do not meet the above criteria, because they provide important information for the adjudication of these events. |
| include urgent<br>outpatient<br>visits. HF<br>hospitalizations<br>should remain | | 5. The subject receives initiation or intensification of treatment specifically for HF, including at least ONE of the following: |
| delineated from | | a. Augmentation in oral diuretic therapy |
| urgent visits. If urgent visits are | | b. Intravenous diuretic or vasoactive agent (eg, inotrope, vasopressor, or vasodilator) |
| included in the HF endpoint, | | c. Mechanical or surgical intervention, including: |
| the number of urgent visits needs to be explicitly | | i.Mechanical circulatory support (eg, intra-aortic balloon pump, ventricular assist device, extracorporeal membrane oxygenation, total artificial heart) |
| presented<br>separately from<br>the | | ii.Mechanical fluid removal (eg, ultrafiltration, hemofiltration, dialysis) |
| hospitalizations. | | An urgent HF visit is defined as an event that meets all of the following: |
| | | 6. The subject has an urgent, unscheduled office/practice or emergency department visit for a primary diagnosis of HF, but not meeting the criteria for a HF hospitalization (i.e. urgent outpatient visit) |
| | | 7. All signs and symptoms for HF hospitalization (ie, symptoms and physical examination findings/laboratory evidence of |

| Event | Mechanism/Classification | Definitions |
|---|---|---|
| | | new or worsening HF, as indicated above) must be met |
| | | 8. The subject receives initiation or intensification of treatment specifically for HF, as detailed in the above section with the exception of oral diuretic therapy, which will not be sufficient. |

<sup>&</sup>lt;sup>a</sup> ACC/AHA 2007 Guidelines for the Management of Patients with Unstable Angina/Non ST- 954 Elevation Myocardial Infarction: Executive Summary. A Report of the American College of 955 Cardiology/American Heart Association Task Force on Practice Guidelines (Writing 956 Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable 957 Angina/Non ST-Elevation Myocardial Infarction): Developed in Collaboration with the 958 American College of Emergency Physicians, the Society for Cardiovascular Angiography 959 and Interventions, and the Society of Thoracic Surgeons: Endorsed by the American 960 Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic 961 Emergency Medicine, Circulation, 2007, 116:803-877.

b The same criteria are used for supplemental leads V7-V9, and for the Cabrera frontal plane lead grouping. Source: "Standardized Definitions for Cardiovascular and Stroke Endpoint Events in Clinical Trials," dated August 20, 2014, and available at the CDISC website (http://www.cdisc.org/system/files/all/standard/Draft%20Definitions%20for%20CDISC%20August%2020,%202014.pdf)

# APPENDIX E. ATORVASTATIN PRESCRIBING INFORMATION

# ATORVASTATIN CALCIUM- atorvastatin calcium trihydrate tablet, film coated Greenstone LLC

\_\_\_\_\_

#### HIGHLIGHTS OF PRESCRIBING INFORMATION

These highlights do not include all the information needed to use atorvastatin calcium tablets safely and effectively. See full prescribing information for atorvastatin calcium tablets.

Atorvastatin Calcium Tablets for oral administration Initial U.S. Approval: 1996

## ----- INDICATIONS AND USAGE

Atorvastatin calcium is an inhibitor of HMG-CoA reductase (statin) indicated as an adjunct therapy to diet to:

- Reduce the risk of MI, stroke, revascularization procedures, and angina in patients without CHD, but with multiple risk factors (1.1).
- Reduce the risk of MI and stroke in patients with type 2 diabetes without CHD, but with multiple risk factors (1.1).
- Reduce the risk of non-fatal MI, fatal and non-fatal stroke, revascularization procedures, hospitalization for CHF, and angina in patients with CHD (1.1).
- Reduce elevated total-C, LDL-C, apo B, and TG levels and increase HDL-C in adult patients with primary hyperlipidemia (heterozygous familial and nonfamilial) and mixed dyslipidemia (1.2).
- Reduce elevated TG in patients with hypertriglyceridemia and primary dysbetalipoproteinemia (1.2).
- Reduce total-C and LDL-C in patients with homozygous familial hypercholesterolemia (HoFH) (1.2).
- Reduce elevated total-C, LDL-C, and apo B levels in boys and postmenarchal girls, 10 to 17 years of age, with heterozygous familial hypercholesterolemia after failing an adequate trial of diet therapy (1.2).

Limitations of Use

Atorvastatin calcium tablets have not been studied in *Fredrickson* Types I and V dyslipidemias.

----- DOSAGE AND ADMINISTRATION -----

Dose range: 10 to 80 mg once daily (2.1).

Recommended start dose: 10 or 20 mg once daily (2.1).

Patients requiring large LDL-C reduction (>45%) may start at 40 mg once daily (2.1).

Pediatric starting dose: 10 mg once daily; maximum recommended dose: 20 mg once daily (2.2).

10, 20, 40, and 80 mg tablets (3).

------CONTRAINDICATIONS

Active liver disease, which may include unexplained persistent elevations in hepatic transaminase levels (4.1).

Women who are pregnant or may become pregnant (4.3). Nursing mothers (4.4).

Hypersensitivity to any component of this medication (4.2).

----- WARNINGS AND PRECAUTIONS -----

Skeletal muscle effects (e.g., myopathy and rhabdomyolysis): Risks increase when higher doses are used concomitantly with cyclosporine and strong CYP3A4 inhibitors (e.g., clarithromycin, itraconazole,

HIV protease inhibitors). Predisposing factors include advanced age (> 65), uncontrolled hypothyroidism, and renal impairment. Rare cases of rhabdomyolysis with acute renal failure secondary to myoglobinuria have been reported. Advise patients to promptly report to their physician unexplained and/or persistent muscle pain, tenderness, or weakness. Atorvastatin therapy should be discontinued if myopathy is diagnosed or suspected (5.1, 8.5).

Liver enzyme abnormalities: Persistent elevations in hepatic transaminases can occur. Check liver enzyme tests before initiating therapy and as clinically indicated thereafter (5.2).

A higher incidence of hemorrhagic stroke was seen in patients without CHD but with stroke or TIA within the previous 6 months in the atorvastatin calcium tablets 80 mg group vs. placebo (5.5).

## -----ADVERSE REACTIONS -----

The most commonly reported adverse reactions (incidence  $\geq 2\%$ ) in patients treated with atorvastatin calcium tablets in placebocontrolled trials regardless of causality were: nasopharyngitis, arthralgia, diarrhea, pain in extremity, and urinary tract infection (6.1).

To report SUSPECTED ADVERSE REACTIONS, contact Greenstone LLC at 1-800-438-1985 or FDA at 1-800-FDA-1088 or www.fda.gov/medwatch.

-----DRUG INTERACTIONS -----

Drug Interactions Associated with Increased Risk of Myopathy/Rhabdomyolysis (2.6, 5.1, 7, 12.3)

| <b>Interacting Agents</b> | Prescribing Recommendations |
|---|---|
| Cyclosporine, HIV protease<br>inhibitors (tipranavir plus<br>ritonavir), hepatitis C protease<br>inhibitor (telaprevir) | Avoid atorvastatin |
| HIV protease inhibitor (lopinavir | Use with caution and lowest |
| plus ritonavir) | dose necessary |
| Clarithromycin, itraconazole,<br>HIV protease inhibitors<br>(saquinavir plus ritonavir,<br>darunavir plus ritonavir,<br>fosamprenavir, fosamprenavir<br>plus ritonavir) | Do not exceed 20 mg atorvastatin daily |
| HIV protease inhibitor<br>(nelfinavir)<br>Hepatitis C protease inhibitor<br>(boceprevir) | Do not exceed 40 mg atorvastatin daily |

- Other Lipid-Lowering Medications: Use with fibrate products or lipid-modifying doses (≥1 g/day) of niacin increases the risk of adverse skeletal muscle effects. Caution should be used when prescribing with atorvastatin calcium tablets (7).
- Digoxin: Patients should be monitored appropriately (7.8).
- Oral Contraceptives: Values for norethindrone and ethinyl estradiol may be increased (7.9).
- Rifampin should be simultaneously co-administered with atorvastatin calcium tablets (7.7).

## ----- USE IN SPECIFIC POPULATIONS

• Hepatic impairment: Plasma concentrations markedly increased in patients with chronic alcoholic liver disease (12.3).

**Revised: 3/2015** 

# FULL PRESCRIBING INFORMATION: CONTENTS\*

### 1 INDICATIONS AND USAGE

- 1.1 Prevention of Cardiovascular Disease
- 1.2 Hyperlipidemia
- 1.3 Limitations of Use

### 2 DOSAGE AND ADMINISTRATION

- 2.1 Hyperlipidemia (Heterozygous Familial and Nonfamilial) and Mixed Dyslipidemia (*Fredrickson* Types IIa and IIb)
- 2.2 Heterozygous Familial Hypercholesterolemia in Pediatric Patients (10–17 years of age)
- 2.3 Homozygous Familial Hypercholesterolemia
- 2.4 Concomitant Lipid-Lowering Therapy
- 2.5 Dosage in Patients With Renal Impairment
- 2.6 Dosage in Patients Taking Cyclosporine, Clarithromycin, Itraconazole, or Certain Protease Inhibitors

# 3 DOSAGE FORMS AND STRENGTHS 4 CONTRAINDICATIONS

- 4.1 Active liver disease, which may include unexplained persistent elevations in hepatic transaminase levels
- 4.2 Hypersensitivity to any component of this medication
- 4.3 Pregnancy
- 4.4 Nursing mothers

### **5 WARNINGS AND PRECAUTIONS**

- 5.1 Skeletal Muscle
- 5.2 Liver Dysfunction
- 5.3 Endocrine Function
- 5.4 CNS Toxicity
- 5.5 Use in Patients with Recent Stroke or TIA

### **6 ADVERSE REACTIONS**

- 6.1 Clinical Trial Adverse Experiences
- 6.2 Postmarketing Experience
- 6.3 Pediatric Patients (ages 10–17 years)

## **7 DRUG INTERACTIONS**

- 7.1 Strong Inhibitors of CYP 3A4
- 7.2 Grapefruit Juice
- 7.3 Cyclosporine
- 7.4 Gemfibrozil
- 7.5 Other Fibrates
- 7.6 Niacin
- 7.7 Rifampin or other Inducers of Cytochrome P450 3A4

- 7.8 Digoxin
- 7.9 Oral Contraceptives
- 7.10 Warfarin
- 7 11 Colchicine

# **8 USE IN SPECIFIC POPULATIONS**

- 8.1 Pregnancy
- 8.3 Nursing Mothers
- 8.4 Pediatric Use
- 8.5 Geriatric Use
- 8.6 Hepatic Impairment
- 10 OVERDOSAGE
- 11 DESCRIPTION

## 12 CLINICAL PHARMACOLOGY

- 12.1 Mechanism of Action
- 12.2 Pharmacodynamics
- 12.3 Pharmacokinetics

## 13 NONCLINICAL TOXICOLOGY

13.1 Carcinogenesis, Mutagenesis, Impairment of Fertility

### 14 CLINICAL STUDIES

- 14.1 Prevention of Cardiovascular Disease
- 14.2 Hyperlipidemia (Heterozygous Familial and Nonfamilial) and Mixed Dyslipidemia (*Fredrickson* Types IIa and IIb)
- 14.3 Hypertriglyceridemia (*Fredrickson* Type IV)
- 14.4 Dysbetalipoproteinemia (*Fredrickson* Type III)
- 14.5 Homozygous Familial Hypercholesterolemia
- 14.6 Heterozygous Familial Hypercholesterolemia in Pediatric Patients

### 15 REFERENCES

# 16 HOW SUPPLIED/STORAGE AND HANDLING

### 17 PATIENT COUNSELING INFORMATION

- 17 1 Muscle Pain
- 17.2 Liver Enzymes
- 17.3 Pregnancy
- 17.4 Breast-feeding
- \* Sections or subsections omitted from the full prescribing information are not listed.

### **FULL PRESCRIBING INFORMATION**

### 1 INDICATIONS AND USAGE

Therapy with lipid-altering agents should be only one component of multiple risk factor intervention in individuals at significantly increased risk for atherosclerotic vascular disease due to hypercholesterolemia. Drug therapy is recommended as an adjunct to diet when the response to a diet restricted in saturated fat and cholesterol and other nonpharmacologic measures alone has been inadequate. In patients with CHD or multiple risk factors for CHD, atorvastatin calcium tablets can be started simultaneously with diet.

### 1.1 Prevention of Cardiovascular Disease

In adult patients without clinically evident coronary heart disease, but with multiple risk factors for coronary heart disease such as age, smoking, hypertension, low HDL-C, or a family history of early coronary heart disease, atorvastatin calcium tablets are indicated to:

- Reduce the risk of myocardial infarction
- Reduce the risk of stroke
- Reduce the risk for revascularization procedures and angina

In patients with type 2 diabetes, and without clinically evident coronary heart disease, but with multiple risk factors for coronary heart disease such as retinopathy, albuminuria, smoking, or hypertension, atorvastatin calcium tablets are indicated to:

- Reduce the risk of myocardial infarction
- Reduce the risk of stroke

In patients with clinically evident coronary heart disease, atorvastatin calcium tablets are indicated to:

- Reduce the risk of non-fatal myocardial infarction
- Reduce the risk of fatal and non-fatal stroke
- Reduce the risk for revascularization procedures
- Reduce the risk of hospitalization for CHF
- Reduce the risk of angina

## 1.2 Hyperlipidemia

Atorvastatin calcium tablets are indicated:

- As an adjunct to diet to reduce elevated total-C, LDL-C, apo B, and TG levels and to increase HDL-C in patients with primary hypercholesterolemia (heterozygous familial and nonfamilial) and mixed dyslipidemia (*Fredrickson* Types IIa and IIb);
- As an adjunct to diet for the treatment of patients with elevated serum TG levels (Fredrickson Type IV);
- For the treatment of patients with primary dysbetalipoproteinemia (Fredrickson Type III) who do not respond adequately to diet;
- To reduce total-C and LDL-C in patients with homozygous familial hypercholesterolemia as an adjunct to other lipid-lowering treatments (e.g., LDL apheresis) or if such treatments are unavailable;
- As an adjunct to diet to reduce total-C, LDL-C, and apo B levels in boys and postmenarchal girls, 10 to 17 years of age, with heterozygous familial hypercholesterolemia if after an adequate trial of diet therapy the following findings are present:
  - a. LDL-C remains ≥ 190 mg/dL or
  - b. LDL-C remains ≥ 160 mg/dL and:
  - there is a positive family history of premature cardiovascular disease or
  - two or more other CVD risk factors are present in the pediatric patient

### 1.3 Limitations of Use

Atorvastatin calcium tablets have not been studied in conditions where the major lipoprotein abnormality is elevation of chylomicrons (*Fredrickson* Types I and V).

### 2 DOSAGE AND ADMINISTRATION

# 2.1 Hyperlipidemia (Heterozygous Familial and Nonfamilial) and Mixed Dyslipidemia (Fredrickson Types IIa and IIb)

The recommended starting dose of atorvastatin calcium tablets is 10 or 20 mg once daily. Patients who require a large reduction in LDL-C (more than 45%) may be started at 40 mg once daily. The dosage range of atorvastatin calcium tablets is 10 to 80 mg once daily. Atorvastatin calcium tablets can be administered as a single dose at any time of the day, with or without food. The starting dose and maintenance doses of atorvastatin calcium tablets should be individualized according to patient characteristics such as goal of therapy and response (see current *NCEP Guidelines*). After initiation and/or upon titration of atorvastatin calcium tablets, lipid levels should be analyzed within 2 to 4 weeks and dosage adjusted accordingly.

# 2.2 Heterozygous Familial Hypercholesterolemia in Pediatric Patients (10–17 years of age)

The recommended starting dose of atorvastatin calcium tablets is 10 mg/day; the maximum recommended dose is 20 mg/day (doses greater than 20 mg have not been studied in this patient population). Doses should be individualized according to the recommended goal of therapy [see current *NCEP Pediatric Panel Guidelines*, *Clinical Pharmacology (12)*, and *Indications and Usage (1.2)*]. Adjustments should be made at intervals of 4 weeks or more.

# 2.3 Homozygous Familial Hypercholesterolemia

The dosage of atorvastatin calcium tablets in patients with homozygous FH is 10 to 80 mg daily. Atorvastatin calcium tablets should be used as an adjunct to other lipid-lowering treatments (e.g., LDL apheresis) in these patients or if such treatments are unavailable.

# 2.4 Concomitant Lipid-Lowering Therapy

Atorvastatin calcium tablets may be used with bile acid resins. The combination of HMG-CoA reductase inhibitors (statins) and fibrates should generally be used with caution [see *Warnings and Precautions, Skeletal Muscle (5.1), Drug Interactions (7)*].

## 2.5 Dosage in Patients With Renal Impairment

Renal disease does not affect the plasma concentrations nor LDL-C reduction of atorvastatin calcium tablets; thus, dosage adjustment in patients with renal dysfunction is not necessary [see *Warnings and Precautions, Skeletal Muscle (5.1), Clinical Pharmacology, Pharmacokinetics (12.3)*].

### 2.6 Dosage in Patients Taking Cyclosporine, Clarithromycin, Itraconazole, or Certain Protease Inhibitors

In patients taking cyclosporine or the HIV protease inhibitors (tipranavir plus ritonavir) or the hepatitis C protease inhibitor (telaprevir), therapy with atorvastatin calcium tablets should be avoided. In patients with HIV taking lopinavir plus ritonavir, caution should be used when prescribing atorvastatin calcium tablets and the lowest dose necessary employed. In patients taking clarithromycin, itraconazole, or in patients with HIV taking a combination of saquinavir plus ritonavir, darunavir plus ritonavir, fosamprenavir, or fosamprenavir plus ritonavir, therapy with atorvastatin calcium tablets should be limited to 20 mg, and appropriate clinical assessment is recommended to ensure that the lowest dose necessary of atorvastatin calcium tablets is employed. In patients taking the HIV protease inhibitor nelfinavir or the hepatitis C protease inhibitor boceprevir, therapy with atorvastatin calcium tablets should be limited to 40 mg, and appropriate clinical assessment is recommended to ensure that the lowest dose necessary of atorvastatin calcium tablets is employed [see *Warnings and Precautions, Skeletal Muscle (5.1), Drug Interactions* (7)].

### **3 DOSAGE FORMS AND STRENGTHS**

White, elliptical, film-coated tablets containing 10, 20, 40, and 80 mg atorvastatin calcium.

### 4 CONTRAINDICATIONS

- 4.1 Active liver disease, which may include unexplained persistent elevations in hepatic transaminase levels
- 4.2 Hypersensitivity to any component of this medication

# 4.3 Pregnancy

Women who are pregnant or may become pregnant. Atorvastatin calcium tablets may cause fetal harm when administered to a pregnant woman. Serum cholesterol and triglycerides increase during normal pregnancy, and cholesterol or cholesterol derivatives are essential for fetal development. Atherosclerosis is a chronic process and discontinuation of lipid-lowering drugs during pregnancy should have little impact on the outcome of long-term therapy of primary hypercholesterolemia. There are no adequate and well-controlled studies of atorvastatin calcium tablets use during pregnancy; however in rare reports, congenital anomalies were observed following intrauterine exposure to statins. In rat and rabbit animal reproduction studies, atorvastatin revealed no evidence of teratogenicity. ATORVASTATIN CALCIUM TABLETS SHOULD BE ADMINISTERED TO WOMEN OF CHILDBEARING AGE ONLY WHEN SUCH PATIENTS ARE HIGHLY UNLIKELY TO CONCEIVE AND HAVE BEEN INFORMED OF THE POTENTIAL HAZARDS. If the patient becomes pregnant while taking this drug, atorvastatin calcium tablets should be discontinued immediately and the patient apprised of the potential hazard to the fetus [see *Use in Specific Populations (8.1)*].

## 4.4 Nursing mothers

It is not known whether atorvastatin is excreted into human milk; however a small amount of another drug in this class does pass into breast milk. Because statins have the potential for serious adverse reactions in nursing infants, women who require atorvastatin calcium tablets treatment should not breastfeed their infants [see *Use in Specific Populations* (8.3)].

### **5 WARNINGS AND PRECAUTIONS**

#### **5.1 Skeletal Muscle**

Rare cases of rhabdomyolysis with acute renal failure secondary to myoglobinuria have been reported with atorvastatin calcium tablets and with other drugs in this class. A history of renal impairment may be a risk factor for the development of rhabdomyolysis. Such patients merit closer monitoring for skeletal muscle effects.

Atorvastatin, like other statins, occasionally causes myopathy, defined as muscle aches or muscle weakness in conjunction with increases in creatine phosphokinase (CPK) values >10 times ULN. The concomitant use of higher doses of atorvastatin with certain drugs such as cyclosporine and strong CYP3A4 inhibitors (e.g., clarithromycin, itraconazole, and HIV protease inhibitors) increases the risk of myopathy/rhabdomyolysis.

There have been rare reports of immune-mediated necrotizing myopathy (IMNM), an autoimmune myopathy, associated with statin use. IMNM is characterized by: proximal muscle weakness and elevated serum creatine kinase,

which persist despite discontinuation of statin treatment; muscle biopsy showing necrotizing myopathy without significant inflammation; improvement with immunosuppressive agents.

Myopathy should be considered in any patient with diffuse myalgias, muscle tenderness or weakness, and/or marked elevation of CPK. Patients should be advised to report promptly unexplained muscle pain, tenderness, or weakness, particularly if accompanied by malaise or fever or if muscle signs and symptoms persist after discontinuing atorvastatin calcium tablets. Atorvastatin therapy should be discontinued if markedly elevated CPK levels occur or myopathy is diagnosed or suspected.

The risk of myopathy during treatment with drugs in this class is increased with concurrent administration of cyclosporine, fibric acid derivatives, erythromycin, clarithromycin, the hepatitis C protease inhibitor telaprevir, combinations of HIV protease inhibitors, including saquinavir plus ritonavir, lopinavir plus ritonavir, tipranavir plus ritonavir, darunavir plus ritonavir, fosamprenavir, and fosamprenavir plus ritonavir, niacin, or azole antifungals. Physicians considering combined therapy with atorvastatin and fibric acid derivatives, erythromycin, clarithromycin, a combination of saquinavir plus ritonavir, lopinavir plus ritonavir, darunavir plus ritonavir, fosamprenavir, or fosamprenavir plus ritonavir, azole antifungals, or lipid-modifying doses of niacin should carefully weigh the potential benefits and risks and should carefully monitor patients for any signs or symptoms of muscle pain, tenderness, or weakness, particularly during the initial months of therapy and during any periods of upward dosage titration of either drug. Lower starting and maintenance doses of atorvastatin should be considered when taken concomitantly with the aforementioned drugs (see *Drug Interactions* (7)). Periodic creatine phosphokinase (CPK) determinations may be considered in such situations, but there is no assurance that such monitoring will prevent the occurrence of severe myopathy.

Prescribing recommendations for interacting agents are summarized in Table 1 [see also *Dosage and Administration* (2.6), *Drug Interactions* (7), *Clinical Pharmacology* (12.3)].

Table 1. Drug Interactions Associated with Increased Risk of Myopathy/Rhabdomyolysis

| Interacting Agents | Prescribing Recommendations |
|---|---|
| Cyclosporine, HIV protease inhibitors (tipranavir plus ritonavir), hepatitis C protease inhibitor (telaprevir) | Avoid atorvastatin |
| HIV protease inhibitor (lopinavir plus ritonavir) | Use with caution and lowest dose necessary |
| Clarithromycin, itraconazole, HIV protease inhibitors (saquinavir plus ritonavir*, darunavir plus ritonavir, fosamprenavir, fosamprenavir plus ritonavir) | Do not exceed 20 mg atorvastatin daily |
| HIV protease inhibitor (nelfinavir)<br>Hepatitis C protease inhibitor<br>(boceprevir) | Do not exceed 40 mg atorvastatin daily |

<sup>\*</sup> Use with caution and with the lowest dose necessary (12.3)

Cases of myopathy, including rhabdomyolysis, have been reported with atorvastatin co-administered with colchicine, and caution should be exercised when prescribing atorvastatin with colchicine [see *Drug Interactions* (7.11)].

Atorvastatin therapy should be temporarily withheld or discontinued in any patient with an acute, serious condition suggestive of a myopathy or having a risk factor predisposing to the development of renal failure secondary to rhabdomyolysis (e.g., severe acute infection, hypotension, major surgery, trauma, severe metabolic, endocrine and electrolyte disorders, and uncontrolled seizures).

# **5.2** Liver Dysfunction

Statins, like some other lipid-lowering therapies, have been associated with biochemical abnormalities of liver function. Persistent elevations (>3 times the upper limit of normal [ULN] occurring on 2 or more occasions) in serum transaminases occurred in 0.7% of patients who received atorvastatin calcium tablets in clinical trials. The incidence of these abnormalities was 0.2%, 0.2%, 0.6%, and 2.3% for 10, 20, 40, and 80 mg, respectively.

One patient in clinical trials developed jaundice. Increases in liver function tests (LFT) in other patients were not associated with jaundice or other clinical signs or symptoms. Upon dose reduction, drug interruption, or discontinuation, transaminase levels returned to or near pretreatment levels without sequelae. Eighteen of 30 patients with persistent LFT elevations continued treatment with a reduced dose of atorvastatin calcium tablets.

It is recommended that liver enzyme tests be obtained prior to initiating therapy with atorvastatin calcium tablets and repeated as clinically indicated. There have been rare postmarketing reports of fatal and non-fatal hepatic failure in patients taking statins, including atorvastatin. If serious liver injury with clinical symptoms and/or hyperbilirubinemia or jaundice occurs during treatment with atorvastatin calcium tablets, promptly interrupt therapy. If an alternate etiology is not found, do not restart atorvastatin calcium tablets.

Atorvastatin calcium tablets should be used with caution in patients who consume substantial quantities of alcohol and/or have a history of liver disease. Active liver disease or unexplained persistent transaminase elevations are contraindications to the use of atorvastatin calcium tablets [see *Contraindications (4.1)*].

### **5.3 Endocrine Function**

Increases in HbA1c and fasting serum glucose levels have been reported with HMG-CoA reductase inhibitors, including atorvastatin calcium tablets.

Statins interfere with cholesterol synthesis and theoretically might blunt adrenal and/or gonadal steroid production. Clinical studies have shown that atorvastatin does not reduce basal plasma cortisol concentration or impair adrenal reserve. The effects of statins on male fertility have not been studied in adequate numbers of patients. The effects, if any, on the pituitary-gonadal axis in premenopausal women are unknown. Caution should be exercised if a statin is administered concomitantly with drugs that may decrease the levels or activity of endogenous steroid hormones, such as ketoconazole, spironolactone, and cimetidine.

## **5.4 CNS Toxicity**

Brain hemorrhage was seen in a female dog treated for 3 months at 120 mg/kg/day. Brain hemorrhage and optic nerve vacuolation were seen in another female dog that was sacrificed in moribund condition after 11 weeks of escalating doses up to 280 mg/kg/day. The 120 mg/kg dose resulted in a systemic exposure approximately 16 times the human plasma area-under-the-curve (AUC, 0–24 hours) based on the maximum human dose of 80 mg/day. A single tonic convulsion was seen in each of 2 male dogs (one treated at 10 mg/kg/day and one at 120 mg/kg/day) in a 2-year study. No CNS lesions have been observed in mice after chronic treatment for up to 2 years at doses up to 400 mg/kg/day or in rats at doses up to 100 mg/kg/day. These doses were 6 to 11 times (mouse) and 8 to 16 times (rat) the human AUC (0–24) based on the maximum recommended human dose of 80 mg/day.

CNS vascular lesions, characterized by perivascular hemorrhages, edema, and mononuclear cell infiltration of perivascular spaces, have been observed in dogs treated with other members of this class. A chemically similar drug in this class produced optic nerve degeneration (Wallerian degeneration of retinogeniculate fibers) in clinically normal dogs in a dose-dependent fashion at a dose that produced plasma drug levels about 30 times higher than the mean drug level in humans taking the highest recommended dose.

### 5.5 Use in Patients with Recent Stroke or TIA

In a post-hoc analysis of the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) study where atorvastatin calcium tablets 80 mg vs. placebo was administered in 4,731 subjects without CHD who had a

stroke or TIA within the preceding 6 months, a higher incidence of hemorrhagic stroke was seen in the atorvastatin calcium tablets 80 mg group compared to placebo (55, 2.3% atorvastatin vs. 33, 1.4% placebo; HR: 1.68, 95% CI: 1.09, 2.59; p=0.0168). The incidence of fatal hemorrhagic stroke was similar across treatment groups (17 vs. 18 for the atorvastatin and placebo groups, respectively). The incidence of nonfatal hemorrhagic stroke was significantly higher in the atorvastatin group (38, 1.6%) as compared to the placebo group (16, 0.7%). Some baseline characteristics, including hemorrhagic and lacunar stroke on study entry, were associated with a higher incidence of hemorrhagic stroke in the atorvastatin group [see *Adverse Reactions* (6.1)].

### **6 ADVERSE REACTIONS**

The following serious adverse reactions are discussed in greater detail in other sections of the label:

Rhabdomyolysis and myopathy [see *Warnings and Precautions (5.1)*]

Liver enzyme abnormalities [see *Warnings and Precautions (5.2)*]

# **6.1 Clinical Trial Adverse Experiences**

Because clinical trials are conducted under widely varying conditions, the adverse reaction rates observed in the clinical studies of a drug cannot be directly compared to rates in the clinical trials of another drug and may not reflect the rates observed in clinical practice.

In the atorvastatin calcium tablets placebo-controlled clinical trial database of 16,066 patients (8755 atorvastatin calcium tablets vs. 7311 placebo; age range 10–93 years, 39% women, 91% Caucasians, 3% Blacks, 2% Asians, 4% other) with a median treatment duration of 53 weeks, 9.7% of patients on atorvastatin calcium tablets and 9.5% of the patients on placebo discontinued due to adverse reactions regardless of causality. The five most common adverse reactions in patients treated with atorvastatin calcium tablets that led to treatment discontinuation and occurred at a rate greater than placebo were: myalgia (0.7%), diarrhea (0.5%), nausea (0.4%), alanine aminotransferase increase (0.4%), and hepatic enzyme increase (0.4%).

The most commonly reported adverse reactions (incidence  $\geq 2\%$  and greater than placebo) regardless of causality, in patients treated with atorvastatin calcium tablets in placebo controlled trials (n=8755) were: nasopharyngitis (8.3%), arthralgia (6.9%), diarrhea (6.8%), pain in extremity (6.0%), and urinary tract infection (5.7%).

Table 2 summarizes the frequency of clinical adverse reactions, regardless of causality, reported in  $\geq$  2% and at a rate greater than placebo in patients treated with atorvastatin calcium tablets (n=8755), from seventeen placebo-controlled trials.

Table 2. Clinical adverse reactions occurring in  $\geq 2\%$  in patients treated with any dose of atorvastatin calcium tablets and at an incidence greater than placebo regardless of causality (% of patients).

| Adverse Reaction* | Any dose<br>N=8755 | 10 mg<br>N=3908 | 20 mg<br>N=188 | 40 mg<br>N=604 | 80 mg<br>N=4055 | Placebo<br>N=7311 |
|---|---|---|---|---|---|---|
| Nasopharyngitis | 8.3 | 12.9 | 5.3 | 7.0 | 4.2 | 8.2 |
| Arthralgia | 6.9 | 8.9 | 11.7 | 10.6 | 4.3 | 6.5 |
| Diarrhea | 6.8 | 7.3 | 6.4 | 14.1 | 5.2 | 6.3 |
| Pain in extremity | 6.0 | 8.5 | 3.7 | 9.3 | 3.1 | 5.9 |
| Urinary tract infection | 5.7 | 6.9 | 6.4 | 8.0 | 4.1 | 5.6 |
| Dyspepsia | 4.7 | 5.9 | 3.2 | 6.0 | 3.3 | 4.3 |
| Nausea | 4.0 | 3.7 | 3.7 | 7.1 | 3.8 | 3.5 |
| Musculoskeletal pain | 3.8 | 5.2 | 3.2 | 5.1 | 2.3 | 3.6 |
| Muscle Spasms | 3.6 | 4.6 | 4.8 | 5.1 | 2.4 | 3.0 |

| Myalgia | 3.5 | 3.6 | 5.9 | 8.4 | 2.7 | 3.1 |
|------------------------|-----|-----|-----|-----|-----|-----|
| Insomnia | 3.0 | 2.8 | 1.1 | 5.3 | 2.8 | 2.9 |
| Pharyngolaryngeal pain | 2.3 | 3.9 | 1.6 | 2.8 | 0.7 | 2.1 |

<sup>\*</sup> Adverse Reaction  $\geq 2\%$  in any dose greater than placebo

Other adverse reactions reported in placebo-controlled studies include:

Body as a whole: malaise, pyrexia; Digestive system: abdominal discomfort, eructation, flatulence, hepatitis, cholestasis; Musculoskeletal system: musculoskeletal pain, muscle fatigue, neck pain, joint swelling; Metabolic and nutritional system: transaminases increase, liver function test abnormal, blood alkaline phosphatase increase, creatine phosphokinase increase, hyperglycemia; Nervous system: nightmare; Respiratory system: epistaxis; Skin and appendages: urticaria; Special senses: vision blurred, tinnitus; Urogenital system: white blood cells urine positive.

## Anglo-Scandinavian Cardiac Outcomes Trial (ASCOT)

In ASCOT [see *Clinical Studies (14.1)*] involving 10,305 participants (age range 40–80 years, 19% women; 94.6% Caucasians, 2.6% Africans, 1.5% South Asians, 1.3% mixed/other) treated with atorvastatin calcium tablets 10 mg daily (n=5,168) or placebo (n=5,137), the safety and tolerability profile of the group treated with atorvastatin calcium tablets was comparable to that of the group treated with placebo during a median of 3.3 years of follow-up.

## Collaborative Atorvastatin Diabetes Study (CARDS)

In CARDS [see *Clinical Studies (14.1)*] involving 2,838 subjects (age range 39–77 years, 32% women; 94.3% Caucasians, 2.4% South Asians, 2.3% Afro-Caribbean, 1.0% other) with type 2 diabetes treated with atorvastatin calcium tablets 10 mg daily (n=1,428) or placebo (n=1,410), there was no difference in the overall frequency of adverse reactions or serious adverse reactions between the treatment groups during a median follow-up of 3.9 years. No cases of rhabdomyolysis were reported.

### *Treating to New Targets Study (TNT)*

In TNT [see *Clinical Studies (14.1)*] involving 10,001 subjects (age range 29–78 years, 19% women; 94.1% Caucasians, 2.9% Blacks, 1.0% Asians, 2.0% other) with clinically evident CHD treated with atorvastatin calcium tablets 10 mg daily (n=5006) or atorvastatin calcium tablets 80 mg daily (n=4995), there were more serious adverse reactions and discontinuations due to adverse reactions in the high-dose atorvastatin group (92, 1.8%; 497, 9.9%, respectively) as compared to the low-dose group (69, 1.4%; 404, 8.1%, respectively) during a median follow-up of 4.9 years. Persistent transaminase elevations ( $\geq$ 3 × ULN twice within 4–10 days) occurred in 62 (1.3%) individuals with atorvastatin 80 mg and in nine (0.2%) individuals with atorvastatin 10 mg. Elevations of CK ( $\geq$  10 × ULN) were low overall, but were higher in the high-dose atorvastatin treatment group (13, 0.3%) compared to the low-dose atorvastatin group (6, 0.1%).

## Incremental Decrease in Endpoints through Aggressive Lipid Lowering Study (IDEAL)

In IDEAL [see *Clinical Studies (14.1)*] involving 8,888 subjects (age range 26–80 years, 19% women; 99.3% Caucasians, 0.4% Asians, 0.3% Blacks, 0.04% other) treated with atorvastatin calcium tablets 80 mg/day (n=4439) or simvastatin 20–40 mg daily (n=4449), there was no difference in the overall frequency of adverse reactions or serious adverse reactions between the treatment groups during a median follow-up of 4.8 years.

## Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL)

In SPARCL involving 4731 subjects (age range 21–92 years, 40% women; 93.3% Caucasians, 3.0% Blacks, 0.6% Asians, 3.1% other) without clinically evident CHD but with a stroke or transient ischemic attack (TIA) within the previous 6 months treated with atorvastatin calcium tablets 80 mg (n=2365) or placebo (n=2366) for a median follow-up of 4.9 years, there was a higher incidence of persistent hepatic transaminase elevations (≥ 3 × ULN twice
within 4–10 days) in the atorvastatin group (0.9%) compared to placebo (0.1%). Elevations of CK (>10 × ULN) were rare, but were higher in the atorvastatin group (0.1%) compared to placebo (0.0%). Diabetes was reported as an adverse reaction in 144 subjects (6.1%) in the atorvastatin group and 89 subjects (3.8%) in the placebo group [see *Warnings and Precautions (5.5)*].

In a post-hoc analysis, atorvastatin calcium tablets 80 mg reduced the incidence of ischemic stroke (218/2365, 9.2% vs. 274/2366, 11.6%) and increased the incidence of hemorrhagic stroke (55/2365, 2.3% vs. 33/2366, 1.4%) compared to placebo. The incidence of fatal hemorrhagic stroke was similar between groups (17 atorvastatin calcium tablets vs. 18 placebo). The incidence of non-fatal hemorrhagic strokes was significantly greater in the atorvastatin group (38 non-fatal hemorrhagic strokes) as compared to the placebo group (16 non-fatal hemorrhagic strokes). Subjects who entered the study with a hemorrhagic stroke appeared to be at increased risk for hemorrhagic stroke [7 (16%) atorvastatin calcium tablets vs. 2 (4%) placebo].

There were no significant differences between the treatment groups for all-cause mortality: 216 (9.1%) in the atorvastatin calcium tablets 80 mg/day group vs. 211 (8.9%) in the placebo group. The proportions of subjects who experienced cardiovascular death were numerically smaller in the atorvastatin calcium tablets 80 mg group (3.3%) than in the placebo group (4.1%). The proportions of subjects who experienced non-cardiovascular death were numerically larger in the atorvastatin calcium tablets 80 mg group (5.0%) than in the placebo group (4.0%).

# **6.2 Postmarketing Experience**

The following adverse reactions have been identified during postapproval use of atorvastatin calcium tablets. Because these reactions are reported voluntarily from a population of uncertain size, it is not always possible to reliably estimate their frequency or establish a causal relationship to drug exposure.

Adverse reactions associated with atorvastatin therapy reported since market introduction, that are not listed above, regardless of causality assessment, include the following: anaphylaxis, angioneurotic edema, bullous rashes (including erythema multiforme, Stevens-Johnson syndrome, and toxic epidermal necrolysis), rhabdomyolysis, myositis, fatigue, tendon rupture, fatal and non-fatal hepatic failure, dizziness, depression, peripheral neuropathy, and pancreatitis.

There have been rare reports of immune-mediated necrotizing myopathy associated with statin use [see *Warnings and Precautions (5.1)*].

There have been rare postmarketing reports of cognitive impairment (e.g., memory loss, forgetfulness, amnesia, memory impairment, confusion) associated with statin use. These cognitive issues have been reported for all statins. The reports are generally nonserious, and reversible upon statin discontinuation, with variable times to symptom onset (1 day to years) and symptom resolution (median of 3 weeks).

# 6.3 Pediatric Patients (ages 10–17 years)

In a 26-week controlled study in boys and postmenarchal girls (n=140, 31% female; 92% Caucasians, 1.6% Blacks, 1.6% Asians, 4.8% other), the safety and tolerability profile of atorvastatin calcium tablets 10 to 20 mg daily was generally similar to that of placebo [see *Clinical Studies (14.6)* and *Use in Special Populations, Pediatric Use (8.4)*].

# 7 DRUG INTERACTIONS

The risk of myopathy during treatment with statins is increased with concurrent administration of fibric acid derivatives, lipid-modifying doses of niacin, cyclosporine, or strong CYP 3A4 inhibitors (e.g., clarithromycin, HIV protease inhibitors, and itraconazole) [see *Warnings and Precautions, Skeletal Muscle (5.1)* and *Clinical Pharmacology (12.3)*].

### 7.1 Strong Inhibitors of CYP 3A4

Atorvastatin is metabolized by cytochrome P450 3A4. Concomitant administration of atorvastatin calcium tablets with strong inhibitors of CYP 3A4 can lead to increases in plasma concentrations of atorvastatin. The extent of interaction and potentiation of effects depend on the variability of effect on CYP 3A4.

Clarithromycin: Atorvastatin AUC was significantly increased with concomitant administration of atorvastatin calcium tablets 80 mg with clarithromycin (500 mg twice daily) compared to that of atorvastatin calcium tablets alone [see *Clinical Pharmacology (12.3)*]. Therefore, in patients taking clarithromycin, caution should be used when the atorvastatin dose exceeds 20 mg [see *Warnings and Precautions, Skeletal Muscle (5.1)* and *Dosage and Administration (2.6)*].

Combination of Protease Inhibitors: Atorvastatin AUC was significantly increased with concomitant administration of atorvastatin calcium tablets with several combinations of HIV protease inhibitors, as well as with the hepatitis C protease inhibitor telaprevir, compared to that of atorvastatin calcium tablets alone [see *Clinical Pharmacology (12.3)*]. Therefore, in patients taking the HIV protease inhibitor tipranavir plus ritonavir, or the hepatitis C protease inhibitor telaprevir, concomitant use of atorvastatin calcium tablets should be avoided. In patients taking the HIV protease inhibitor lopinavir plus ritonavir, caution should be used when prescribing atorvastatin calcium tablets and the lowest dose necessary should be used. In patients taking the HIV protease inhibitors saquinavir plus ritonavir, darunavir plus ritonavir, fosamprenavir, or fosamprenavir plus ritonavir, the dose of atorvastatin calcium tablets should not exceed 20 mg and should be used with caution [see *Warnings and Precautions, Skeletal Muscle (5.1)* and *Dosage and Administration (2.6)*]. In patients taking the HIV protease inhibitor nelfinavir or the hepatitis C protease inhibitor boceprevir, the dose of atorvastatin calcium tablets should not exceed 40 mg and close clinical monitoring is recommended.

**Itraconazole:** Atorvastatin AUC was significantly increased with concomitant administration of atorvastatin calcium tablets 40 mg and itraconazole 200 mg [see *Clinical Pharmacology (12.3)*]. Therefore, in patients taking itraconazole, caution should be used when the atorvastatin dose exceeds 20 mg [see *Warnings and Precautions*, *Skeletal Muscle (5.1)* and *Dosage and Administration (2.6)*].

# 7.2 Grapefruit Juice

Contains one or more components that inhibit CYP 3A4 and can increase plasma concentrations of atorvastatin, especially with excessive grapefruit juice consumption (>1.2 liters per day).

# 7.3 Cyclosporine

Atorvastatin and atorvastatin-metabolites are substrates of the OATP1B1 transporter. Inhibitors of the OATP1B1 (e.g., cyclosporine) can increase the bioavailability of atorvastatin. Atorvastatin AUC was significantly increased with concomitant administration of atorvastatin calcium tablets 10 mg and cyclosporine 5.2 mg/kg/day compared to that of atorvastatin calcium tablets alone [see *Clinical Pharmacology (12.3)*]. The co-administration of atorvastatin calcium tablets with cyclosporine should be avoided [see *Warnings and Precautions, Skeletal Muscle (5.1)*].

### 7.4 Gemfibrozil

Due to an increased risk of myopathy/rhabdomyolysis when HMG-CoA reductase inhibitors are co-administered with gemfibrozil, concomitant administration of atorvastatin calcium tablets with gemfibrozil should be avoided [see *Warnings and Precautions (5.1)*].

### 7.5 Other Fibrates

Because it is known that the risk of myopathy during treatment with HMG-CoA reductase inhibitors is increased with concurrent administration of other fibrates, atorvastatin calcium tablets should be administered with caution when

used concomitantly with other fibrates [see *Warnings and Precautions (5.1)*].

### 7.6 Niacin

The risk of skeletal muscle effects may be enhanced when atorvastatin calcium tablets are used in combination with niacin; a reduction in atorvastatin calcium tablets dosage should be considered in this setting [see *Warnings and Precautions (5.1)*].

# 7.7 Rifampin or other Inducers of Cytochrome P450 3A4

Concomitant administration of atorvastatin calcium tablets with inducers of cytochrome P450 3A4 (e.g., efavirenz, rifampin) can lead to variable reductions in plasma concentrations of atorvastatin. Due to the dual interaction mechanism of rifampin, simultaneous co-administration of atorvastatin calcium tablets with rifampin is recommended, as delayed administration of atorvastatin after administration of rifampin has been associated with a significant reduction in atorvastatin plasma concentrations.

# 7.8 Digoxin

When multiple doses of atorvastatin calcium tablets and digoxin were coadministered, steady state plasma digoxin concentrations increased by approximately 20%. Patients taking digoxin should be monitored appropriately.

# 7.9 Oral Contraceptives

Co-administration of atorvastatin calcium tablets and an oral contraceptive increased AUC values for norethindrone and ethinyl estradiol [see *Clinical Pharmacology (12.3)*]. These increases should be considered when selecting an oral contraceptive for a woman taking atorvastatin.

### 7.10 Warfarin

Atorvastatin calcium tablets had no clinically significant effect on prothrombin time when administered to patients receiving chronic warfarin treatment.

#### 7.11 Colchicine

Cases of myopathy, including rhabdomyolysis, have been reported with atorvastatin co-administered with colchicine, and caution should be exercised when prescribing atorvastatin with colchicine.

### **8 USE IN SPECIFIC POPULATIONS**

### 8.1 Pregnancy

# Pregnancy Category X

Atorvastatin calcium tablets are contraindicated in women who are or may become pregnant. Serum cholesterol and triglycerides increase during normal pregnancy. Lipid lowering drugs offer no benefit during pregnancy because cholesterol and cholesterol derivatives are needed for normal fetal development. Atherosclerosis is a chronic process, and discontinuation of lipid-lowering drugs during pregnancy should have little impact on long-term outcomes of primary hypercholesterolemia therapy.

There are no adequate and well-controlled studies of atorvastatin use during pregnancy. There have been rare reports

of congenital anomalies following intrauterine exposure to statins. In a review of about 100 prospectively followed pregnancies in women exposed to other statins, the incidences of congenital anomalies, spontaneous abortions, and fetal deaths/stillbirths did not exceed the rate expected in the general population. However, this study was only able to exclude a three-to-four-fold increased risk of congenital anomalies over background incidence. In 89% of these cases, drug treatment started before pregnancy and stopped during the first trimester when pregnancy was identified.

Atorvastatin crosses the rat placenta and reaches a level in fetal liver equivalent to that of maternal plasma. Atorvastatin was not teratogenic in rats at doses up to 300 mg/kg/day or in rabbits at doses up to 100 mg/kg/day. These doses resulted in multiples of about 30 times (rat) or 20 times (rabbit) the human exposure based on surface area (mg/m²) [see *Contraindications, Pregnancy (4.3)*].

In a study in rats given 20, 100, or 225 mg/kg/day, from gestation day 7 through to lactation day 21 (weaning), there was decreased pup survival at birth, neonate, weaning, and maturity in pups of mothers dosed with 225 mg/kg/day. Body weight was decreased on days 4 and 21 in pups of mothers dosed at 100 mg/kg/day; pup body weight was decreased at birth and at days 4, 21, and 91 at 225 mg/kg/day. Pup development was delayed (rotorod performance at 100 mg/kg/day and acoustic startle at 225 mg/kg/day; pinnae detachment and eye-opening at 225 mg/kg/day). These doses correspond to 6 times (100 mg/kg) and 22 times (225 mg/kg) the human AUC at 80 mg/day.

Statins may cause fetal harm when administered to a pregnant woman. Atorvastatin calcium tablets should be administered to women of childbearing potential only when such patients are highly unlikely to conceive and have been informed of the potential hazards. If the woman becomes pregnant while taking atorvastatin, it should be discontinued immediately and the patient advised again as to the potential hazards to the fetus and the lack of known clinical benefit with continued use during pregnancy.

# **8.3 Nursing Mothers**

It is not known whether atorvastatin is excreted in human milk, but a small amount of another drug in this class does pass into breast milk. Nursing rat pups had plasma and liver drug levels of 50% and 40%, respectively, of that in their mother's milk. Animal breast milk drug levels may not accurately reflect human breast milk levels. Because another drug in this class passes into human milk and because statins have a potential to cause serious adverse reactions in nursing infants, women requiring atorvastatin treatment should be advised not to nurse their infants [see *Contraindications (4)*].

### 8.4 Pediatric Use

Safety and effectiveness in patients 10–17 years of age with heterozygous familial hypercholesterolemia have been evaluated in a controlled clinical trial of 6 months' duration in adolescent boys and postmenarchal girls. Patients treated with atorvastatin calcium tablets had an adverse experience profile generally similar to that of patients treated with placebo. The most common adverse experiences observed in both groups, regardless of causality assessment, were infections. **Doses greater than 20 mg have not been studied in this patient population.** In this limited controlled study, there was no significant effect on growth or sexual maturation in boys or on menstrual cycle length in girls [see *Clinical Studies (14.6); Adverse Reactions, Pediatric Patients (ages 10–17 years) (6.3)*; and *Dosage and Administration, Heterozygous Familial Hypercholesterolemia in Pediatric Patients (10–17 years of age) (2.2)*]. Adolescent females should be counseled on appropriate contraceptive methods while on atorvastatin therapy [see *Contraindications, Pregnancy (4.3)* and *Use in Specific Populations, Pregnancy (8.1)*]. **Atorvastatin calcium tablets have not been studied in controlled clinical trials involving pre-pubertal patients or patients younger than 10 years of age.** 

Clinical efficacy with doses up to 80 mg/day for 1 year have been evaluated in an uncontrolled study of patients with homozygous FH including 8 pediatric patients [see *Clinical Studies, Homozygous Familial Hypercholesterolemia* (14.5)].

### 8.5 Geriatric Use

Of the 39,828 patients who received atorvastatin calcium tablets in clinical studies, 15,813 (40%) were ≥65 years old

and 2,800 (7%) were  $\geq$ 75 years old. No overall differences in safety or effectiveness were observed between these subjects and younger subjects, and other reported clinical experience has not identified differences in responses between the elderly and younger patients, but greater sensitivity of some older adults cannot be ruled out. Since advanced age ( $\geq$ 65 years) is a predisposing factor for myopathy, atorvastatin should be prescribed with caution in the elderly.

# 8.6 Hepatic Impairment

Atorvastatin calcium tablets are contraindicated in patients with active liver disease which may include unexplained persistent elevations in hepatic transaminase levels [see *Contraindications (4)* and *Pharmacokinetics (12.3)*].

# 10 OVERDOSAGE

There is no specific treatment for atorvastatin overdosage. In the event of an overdose, the patient should be treated symptomatically, and supportive measures instituted as required. Due to extensive drug binding to plasma proteins, hemodialysis is not expected to significantly enhance atorvastatin clearance.

# 11 DESCRIPTION

Atorvastatin calcium is a synthetic lipid-lowering agent. Atorvastatin is an inhibitor of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase. This enzyme catalyzes the conversion of HMG-CoA to mevalonate, an early and rate-limiting step in cholesterol biosynthesis.

Atorvastatin calcium is  $[R-(R^*, R^*)]-2-(4-fluorophenyl)-\beta$ ,  $\delta$ -dihydroxy-5-(1-methylethyl)-3-phenyl-4-[(phenylamino)carbonyl]-1H-pyrrole-1-heptanoic acid, calcium salt (2:1) trihydrate. The empirical formula of atorvastatin calcium is  $(C_{33}H_{34}FN_2O_5)_2Ca \cdot 3H_2O$  and its molecular weight is 1209.42. Its structural formula is:

Atorvastatin calcium is a white to off-white crystalline powder that is insoluble in aqueous solutions of pH 4 and below. Atorvastatin calcium is very slightly soluble in distilled water, pH 7.4 phosphate buffer, and acetonitrile; slightly soluble in ethanol; and freely soluble in methanol.

Atorvastatin calcium tablets for oral administration contain 10, 20, 40, or 80 mg atorvastatin and the following inactive ingredients: calcium carbonate, USP; candelilla wax, FCC; croscarmellose sodium, NF; hydroxypropyl cellulose, NF; lactose monohydrate, NF; magnesium stearate, NF; microcrystalline cellulose, NF; Opadry White YS-1-7040 (hypromellose, polyethylene glycol, talc, titanium dioxide); polysorbate 80, NF; simethicone emulsion.

### 12 CLINICAL PHARMACOLOGY

# 12.1 Mechanism of Action

Atorvastatin calcium is a selective, competitive inhibitor of HMG-CoA reductase, the rate-limiting enzyme that

converts 3-hydroxy-3-methylglutaryl-coenzyme A to mevalonate, a precursor of sterols, including cholesterol. Cholesterol and triglycerides circulate in the bloodstream as part of lipoprotein complexes. With ultracentrifugation, these complexes separate into HDL (high-density lipoprotein), IDL (intermediate-density lipoprotein), LDL (low-density lipoprotein), and VLDL (very-low-density lipoprotein) fractions. Triglycerides (TG) and cholesterol in the liver are incorporated into VLDL and released into the plasma for delivery to peripheral tissues. LDL is formed from VLDL and is catabolized primarily through the high-affinity LDL receptor. Clinical and pathologic studies show that elevated plasma levels of total cholesterol (total-C), LDL-cholesterol (LDL-C), and apolipoprotein B (apo B) promote human atherosclerosis and are risk factors for developing cardiovascular disease, while increased levels of HDL-C are associated with a decreased cardiovascular risk.

In animal models, atorvastatin lowers plasma cholesterol and lipoprotein levels by inhibiting HMG-CoA reductase and cholesterol synthesis in the liver and by increasing the number of hepatic LDL receptors on the cell surface to enhance uptake and catabolism of LDL; atorvastatin also reduces LDL production and the number of LDL particles. Atorvastatin reduces LDL-C in some patients with homozygous familial hypercholesterolemia (FH), a population that rarely responds to other lipid-lowering medication(s).

A variety of clinical studies have demonstrated that elevated levels of total-C, LDL-C, and apo B (a membrane complex for LDL-C) promote human atherosclerosis. Similarly, decreased levels of HDL-C (and its transport complex, apo A) are associated with the development of atherosclerosis. Epidemiologic investigations have established that cardiovascular morbidity and mortality vary directly with the level of total-C and LDL-C, and inversely with the level of HDL-C.

Atorvastatin reduces total-C, LDL-C, and apo B in patients with homozygous and heterozygous FH, nonfamilial forms of hypercholesterolemia, and mixed dyslipidemia. Atorvastatin also reduces VLDL-C and TG and produces variable increases in HDL-C and apolipoprotein A-1. Atorvastatin reduces total-C, LDL-C, VLDL-C, apo B, TG, and non-HDL-C, and increases HDL-C in patients with isolated hypertriglyceridemia. Atorvastatin reduces intermediate density lipoprotein cholesterol (IDL-C) in patients with dysbetalipoproteinemia.

Like LDL, cholesterol-enriched triglyceride-rich lipoproteins, including VLDL, intermediate density lipoprotein (IDL), and remnants, can also promote atherosclerosis. Elevated plasma triglycerides are frequently found in a triad with low HDL-C levels and small LDL particles, as well as in association with non-lipid metabolic risk factors for coronary heart disease. As such, total plasma TG has not consistently been shown to be an independent risk factor for CHD. Furthermore, the independent effect of raising HDL or lowering TG on the risk of coronary and cardiovascular morbidity and mortality has not been determined.

# 12.2 Pharmacodynamics

Atorvastatin calcium, as well as some of its metabolites, is pharmacologically active in humans. The liver is the primary site of action and the principal site of cholesterol synthesis and LDL clearance. Drug dosage, rather than systemic drug concentration, correlates better with LDL-C reduction. Individualization of drug dosage should be based on therapeutic response [see *Dosage and Administration (2)*].

### 12.3 Pharmacokinetics

Absorption: Atorvastatin calcium tablets are rapidly absorbed after oral administration; maximum plasma concentrations occur within 1 to 2 hours. Extent of absorption increases in proportion to atorvastatin calcium dose. The absolute bioavailability of atorvastatin (parent drug) is approximately 14% and the systemic availability of HMG-CoA reductase inhibitory activity is approximately 30%. The low systemic availability is attributed to presystemic clearance in gastrointestinal mucosa and/or hepatic first-pass metabolism. Although food decreases the rate and extent of drug absorption by approximately 25% and 9%, respectively, as assessed by Cmax and AUC, LDL-C reduction is similar whether atorvastatin calcium tablets are given with or without food. Plasma atorvastatin concentrations are lower (approximately 30% for Cmax and AUC) following evening drug administration compared with morning. However, LDL-C reduction is the same regardless of the time of day of drug administration [see *Dosage and Administration (2)*].

**Distribution:** Mean volume of distribution of atorvastatin is approximately 381 liters. Atorvastatin is ≥98% bound to plasma proteins. A blood/plasma ratio of approximately 0.25 indicates poor drug penetration into red blood cells. Based on observations in rats, atorvastatin is likely to be secreted in human milk [see *Contraindications, Nursing Mothers (4.4)* and *Use in Specific Populations, Nursing Mothers (8.3)*].

**Metabolism:** Atorvastatin is extensively metabolized to ortho- and parahydroxylated derivatives and various beta-oxidation products. *In vitro* inhibition of HMG-CoA reductase by ortho- and parahydroxylated metabolites is equivalent to that of atorvastatin. Approximately 70% of circulating inhibitory activity for HMG-CoA reductase is attributed to active metabolites. *In vitro* studies suggest the importance of atorvastatin metabolism by cytochrome P450 3A4, consistent with increased plasma concentrations of atorvastatin in humans following co-administration with erythromycin, a known inhibitor of this isozyme [see *Drug Interactions (7.1)*]. In animals, the ortho-hydroxy metabolite undergoes further glucuronidation.

**Excretion:** Atorvastatin and its metabolites are eliminated primarily in bile following hepatic and/or extra-hepatic metabolism; however, the drug does not appear to undergo enterohepatic recirculation. Mean plasma elimination half-life of atorvastatin in humans is approximately 14 hours, but the half-life of inhibitory activity for HMG-CoA reductase is 20 to 30 hours due to the contribution of active metabolites. Less than 2% of a dose of atorvastatin calcium tablets is recovered in urine following oral administration.

# **Specific Populations**

**Geriatric:** Plasma concentrations of atorvastatin are higher (approximately 40% for Cmax and 30% for AUC) in healthy elderly subjects (age ≥65 years) than in young adults. Clinical data suggest a greater degree of LDL-lowering at any dose of drug in the elderly patient population compared to younger adults [see *Use in Specific Populations*, *Geriatric Use (8.5)*].

**Pediatric:** Pharmacokinetic data in the pediatric population are not available.

**Gender:** Plasma concentrations of atorvastatin in women differ from those in men (approximately 20% higher for Cmax and 10% lower for AUC); however, there is no clinically significant difference in LDL-C reduction with atorvastatin between men and women.

**Renal Impairment:** Renal disease has no influence on the plasma concentrations or LDL-C reduction of atorvastatin; thus, dose adjustment in patients with renal dysfunction is not necessary [see *Dosage and Administration, Dosage in Patients with Renal Impairment (2.5), Warnings and Precautions, Skeletal Muscle (5.1)].* 

**Hemodialysis:** While studies have not been conducted in patients with end-stage renal disease, hemodialysis is not expected to significantly enhance clearance of atorvastatin since the drug is extensively bound to plasma proteins.

**Hepatic Impairment:** In patients with chronic alcoholic liver disease, plasma concentrations of atorvastatin are markedly increased. Cmax and AUC are each 4-fold greater in patients with Childs-Pugh A disease. Cmax and AUC are approximately 16-fold and 11-fold increased, respectively, in patients with Childs-Pugh B disease [see *Contraindications (4.1)*].

TABLE 3. Effect of Co-administered Drugs on the Pharmacokinetics of Atorvastatin

| Co-administered drug and dosing regimen | Atorvastatin | |
|-----------------------------------------|--------------|-----------|
| | | Change in |

| | Dose (mg) | Change in AUC* | Cmax* |
|---|---|---|---|
| †Cyclosporine 5.2 mg/kg/day, stable dose | 10 mg QD for 28 days | ↑ 8.7 fold | ↑10.7 fold |
| †Tipranavir 500 mg BID/ritonavir 200 mg BID, 7 days | 10 mg, SD | ↑ 9.4 fold | ↑ 8.6 fold |
| <sup>†</sup> Telaprevir 750 mg q8h, 10 days | 20 mg, SD | ↑ 7.88 fold | ↑ 10.6 fold |
| †,‡Saquinavir 400 mg BID/ ritonavir 400 mg<br>BID, 15 days | 40 mg QD for 4 days | ↑ 3.9 fold | ↑ 4.3 fold |
| <sup>†</sup> Clarithromycin 500 mg BID, 9 days | 80 mg QD for 8 days | ↑ 4.4 fold | ↑ 5.4 fold |
| †Darunavir 300 mg BID/ritonavir 100 mg BID, 9 days | 10 mg QD for 4 days | ↑ 3.4 fold | ↑ 2.25 fold |
| †Itraconazole 200 mg QD, 4 days | 40 mg SD | ↑ 3.3 fold | ↑ 20% |
| †Fosamprenavir 700 mg BID/ritonavir 100 mg BID, 14 days | 10 mg QD for 4 days | ↑ 2.53 fold | ↑ 2.84 fold |
| †Fosamprenavir 1400 mg BID, 14 days | 10 mg QD for 4 days | ↑ 2.3 fold | ↑ 4.04 fold |
| <sup>†</sup> Nelfinavir 1250 mg BID, 14 days | 10 mg QD for 28 days | ↑ 74% | ↑ 2.2 fold |
| <sup>†</sup> Grapefruit Juice, 240 mL QD <sup>§</sup> | 40 mg, SD | ↑ 37% | ↑ 16% |
| Diltiazem 240 mg QD, 28 days | 40 mg, SD | ↑ 51% | No change |
| Erythromycin 500 mg QID, 7 days | 10 mg, SD | ↑ 33% | ↑ 38% |
| Amlodipine 10 mg, single dose | 80 mg, SD | ↑ 15% | ↓ 12 % |
| Cimetidine 300 mg QID, 2 weeks | 10 mg QD for 2 weeks | ↓ Less than 1% | ↓ 11% |
| Colestipol 10 mg BID, 28 weeks | 40 mg QD for 28 weeks | Not determined | ↓ 26%¶ |
| Maalox TC® 30 mL QD, 17 days | 10 mg QD for 15 days | ↓ 33% | ↓ 34% |
| Efavirenz 600 mg QD, 14 days | 10 mg for 3 days | ↓ 41% | ↓ 1% |
| †Rifampin 600 mg QD, 7 days (co-administered) | 40 mg SD | ↑ 30% | ↑ 2.7 fold |
| †Rifampin 600 mg QD, 5 days (doses separated) | 40 mg SD | ↓ 80% | ↓ 40% |
| †Gemfibrozil 600mg BID, 7 days | 40mg SD | ↑ 35% | ↓ Less than 1% |
| †Fenofibrate 160mg QD, 7 days | 40mg SD | ↑ 3% | ↑ 2% |
| Boceprevir 800 mg TID, 7 days | 40 mg SD | ↑2.30 fold | ↑2.66 fold |

<sup>\*</sup> Data given as x-fold change represent a simple ratio between co-administration and atorvastatin alone (i.e., 1-fold = no change). Data given as % change represent % difference relative to atorvastatin alone (i.e., 0% = no change).

TABLE 4. Effect of Atorvastatin on the Pharmacokinetics of Co-administered Drugs

| Atorvastatin | Co-administer | red drug and dosing r | egimen |
|--------------|---------------|-----------------------|--------|

<sup>†</sup> See Sections 5.1 and 7 for clinical significance.

The dose of saquinavir plus ritonavir in this study is not the clinically used dose. The increase in atorvastatin exposure when used clinically is likely to be higher than what was observed in this study. Therefore, caution should be applied and the lowest dose necessary should be used.

<sup>§</sup> Greater increases in AUC (up to 2.5 fold) and/or Cmax (up to 71%) have been reported with excessive grapefruit consumption (≥ 750 mL − 1.2 liters per day).

Single sample taken 8–16 h post dose.

<sup>#</sup> Due to the dual interaction mechanism of rifampin, simultaneous co-administration of atorvastatin with rifampin is recommended, as delayed administration of atorvastatin after administration of rifampin has been associated with a significant reduction in atorvastatin plasma concentrations.

| | Drug/Dose (mg) | Change in AUC | Change in Cmax |
|---|---|---|---|
| 80 mg QD for 15 days | Antipyrine, 600 mg SD | ↑ 3% | ↓ 11% |
| 80 mg QD for 14 days | * Digoxin 0.25 mg QD, 20 days | ↑ 15% | ↑ 20 % |
| 40 mg QD for 22 days | Oral contraceptive QD, 2 months | | |
| | - norethindrone 1mg<br>- ethinyl estradiol 35μg | ↑ 28%<br>↑ 19% | ↑ 23%<br>↑ 30% |
| 10 mg, SD | Tipranavir 500 mg<br>BID/ritonavir 200 mg BID, 7<br>days | | No change |
| 10 mg QD for 4 days | Fosamprenavir 1400 mg BID,<br>14 days | ↓ 27% | ↓ 18% |
| 10 mg QD for 4 days | Fosamprenavir 700 mg<br>BID/ritonavir 100 mg BID,<br>14 days | No change | No change |

<sup>\*</sup> See Section 7 for clinical significance.

### 13 NONCLINICAL TOXICOLOGY

# 13.1 Carcinogenesis, Mutagenesis, Impairment of Fertility

In a 2-year carcinogenicity study in rats at dose levels of 10, 30, and 100 mg/kg/day, 2 rare tumors were found in muscle in high-dose females: in one, there was a rhabdomyosarcoma and, in another, there was a fibrosarcoma. This dose represents a plasma AUC (0–24) value of approximately 16 times the mean human plasma drug exposure after an 80 mg oral dose.

A 2-year carcinogenicity study in mice given 100, 200, or 400 mg/kg/day resulted in a significant increase in liver adenomas in high-dose males and liver carcinomas in high-dose females. These findings occurred at plasma AUC (0–24) values of approximately 6 times the mean human plasma drug exposure after an 80 mg oral dose.

*In vitro*, atorvastatin was not mutagenic or clastogenic in the following tests with and without metabolic activation: the Ames test with *Salmonella typhimurium* and *Escherichia coli*, the HGPRT forward mutation assay in Chinese hamster lung cells, and the chromosomal aberration assay in Chinese hamster lung cells. Atorvastatin was negative in the *in vivo* mouse micronucleus test.

Studies in rats performed at doses up to 175 mg/kg (15 times the human exposure) produced no changes in fertility. There was aplasia and aspermia in the epididymis of 2 of 10 rats treated with 100 mg/kg/day of atorvastatin for 3 months (16 times the human AUC at the 80 mg dose); testis weights were significantly lower at 30 and 100 mg/kg and epididymal weight was lower at 100 mg/kg. Male rats given 100 mg/kg/day for 11 weeks prior to mating had decreased sperm motility, spermatid head concentration, and increased abnormal sperm. Atorvastatin caused no adverse effects on semen parameters, or reproductive organ histopathology in dogs given doses of 10, 40, or 120 mg/kg for two years.

### 14 CLINICAL STUDIES

# 14.1 Prevention of Cardiovascular Disease

In the Anglo-Scandinavian Cardiac Outcomes Trial (ASCOT), the effect of atorvastatin on fatal and non-fatal

coronary heart disease was assessed in 10,305 hypertensive patients 40–80 years of age (mean of 63 years), without a previous myocardial infarction and with TC levels ≤251 mg/dL (6.5 mmol/L). Additionally, all patients had at least 3 of the following cardiovascular risk factors: male gender (81.1%), age >55 years (84.5%), smoking (33.2%), diabetes (24.3%), history of CHD in a first-degree relative (26%), TC:HDL >6 (14.3%), peripheral vascular disease (5.1%), left ventricular hypertrophy (14.4%), prior cerebrovascular event (9.8%), specific ECG abnormality (14.3%), proteinuria/albuminuria (62.4%). In this double-blind, placebo-controlled study, patients were treated with anti-hypertensive therapy (Goal BP <140/90 mm Hg for non-diabetic patients; <130/80 mm Hg for diabetic patients) and allocated to either atorvastatin calcium tablets 10 mg daily (n=5168) or placebo (n=5137), using a covariate adaptive method which took into account the distribution of nine baseline characteristics of patients already enrolled and minimized the imbalance of those characteristics across the groups. Patients were followed for a median duration of 3.3 years.

The effect of 10 mg/day of atorvastatin calcium tablets on lipid levels was similar to that seen in previous clinical trials.

Atorvastatin significantly reduced the rate of coronary events [either fatal coronary heart disease (46 events in the placebo group vs. 40 events in the atorvastatin calcium tablets group) or non-fatal MI (108 events in the placebo group vs. 60 events in the atorvastatin calcium tablets group)] with a relative risk reduction of 36% [(based on incidences of 1.9% for atorvastatin calcium tablets vs. 3.0% for placebo), p=0.0005 (see Figure 1)]. The risk reduction was consistent regardless of age, smoking status, obesity, or presence of renal dysfunction. The effect of atorvastatin was seen regardless of baseline LDL levels. Due to the small number of events, results for women were inconclusive.

Figure 1: Effect of Atorvastatin 10 mg/day on Cumulative Incidence of Non-Fatal Myocardial Infarction or Coronary Heart Disease Death (in ASCOT-LLA)



Atorvastatin also significantly decreased the relative risk for revascularization procedures by 42%. Although the reduction of fatal and non-fatal strokes did not reach a pre-defined significance level (p=0.01), a favorable trend was observed with a 26% relative risk reduction (incidences of 1.7% for atorvastatin calcium tablets and 2.3% for placebo). There was no significant difference between the treatment groups for death due to cardiovascular causes (p=0.51) or noncardiovascular causes (p=0.17).

In the Collaborative Atorvastatin Diabetes Study (CARDS), the effect of atorvastatin on cardiovascular disease (CVD) endpoints was assessed in 2838 subjects (94% white, 68% male), ages 40–75 with type 2 diabetes based on WHO criteria, without prior history of cardiovascular disease and with LDL  $\leq$  160 mg/dL and TG  $\leq$  600 mg/dL. In addition to diabetes, subjects had 1 or more of the following risk factors: current smoking (23%), hypertension (80%), retinopathy (30%), or microalbuminuria (9%) or macroalbuminuria (3%). No subjects on hemodialysis were

enrolled in the study. In this multicenter, placebo-controlled, double-blind clinical trial, subjects were randomly allocated to either atorvastatin calcium tablets 10 mg daily (1429) or placebo (1411) in a 1:1 ratio and were followed for a median duration of 3.9 years. The primary endpoint was the occurrence of any of the major cardiovascular events: myocardial infarction, acute CHD death, unstable angina, coronary revascularization, or stroke. The primary analysis was the time to first occurrence of the primary endpoint.

Baseline characteristics of subjects were: mean age of 62 years, mean HbA<sub>1c</sub> 7.7%; median LDL-C 120 mg/dL; median TC 207 mg/dL; median TG 151 mg/dL; median HDL-C 52 mg/dL.

The effect of atorvastatin 10 mg/day on lipid levels was similar to that seen in previous clinical trials.

Atorvastatin significantly reduced the rate of major cardiovascular events (primary endpoint events) (83 events in the atorvastatin calcium tablets group vs. 127 events in the placebo group) with a relative risk reduction of 37%, HR 0.63, 95% CI (0.48, 0.83) (p=0.001) (see Figure 2). An effect of atorvastatin calcium tablets was seen regardless of age, sex, or baseline lipid levels.

Atorvastatin significantly reduced the risk of stroke by 48% (21 events in the atorvastatin calcium tablets group vs. 39 events in the placebo group), HR 0.52, 95% CI (0.31, 0.89) (p=0.016) and reduced the risk of MI by 42% (38 events in the atorvastatin calcium tablets group vs. 64 events in the placebo group), HR 0.58, 95.1% CI (0.39, 0.86) (p=0.007). There was no significant difference between the treatment groups for angina, revascularization procedures, and acute CHD death.

There were 61 deaths in the atorvastatin calcium tablets group vs. 82 deaths in the placebo group (HR 0.73, p=0.059).

Figure 2: Effect of Atorvastatin 10 mg/day on Time to Occurrence of Major Cardiovascular Event (myocardial infarction, acute CHD death, unstable angina, coronary revascularization, or stroke) in CARDS



In the Treating to New Targets Study (TNT), the effect of atorvastatin calcium tablets 80 mg/day vs. atorvastatin calcium tablets 10 mg/day on the reduction in cardiovascular events was assessed in 10,001 subjects (94% white, 81% male, 38% ≥65 years) with clinically evident coronary heart disease who had achieved a target LDL-C level <130 mg/dL after completing an 8-week, open-label, run-in period with atorvastatin calcium tablets 10 mg/day. Subjects were randomly assigned to either 10 mg/day or 80 mg/day of atorvastatin calcium tablets and followed for a median duration of 4.9 years. The primary endpoint was the time-to-first occurrence of any of the following major cardiovascular events (MCVE): death due to CHD, non-fatal myocardial infarction, resuscitated cardiac arrest, and fatal and non-fatal stroke. The mean LDL-C, TC, TG, non-HDL, and HDL cholesterol levels at 12 weeks were 73, 145, 128, 98, and 47 mg/dL during treatment with 80 mg of atorvastatin calcium tablets and 99, 177, 152, 129, and 48 mg/dL during treatment with 10 mg of atorvastatin calcium tablets.

Treatment with atorvastatin calcium tablets 80 mg/day significantly reduced the rate of MCVE (434 events in the 80 mg/day group vs. 548 events in the 10 mg/day group) with a relative risk reduction of 22%, HR 0.78, 95% CI (0.69,

0.89), p=0.0002 (see Figure 3 and Table 5). The overall risk reduction was consistent regardless of age ( $<65, \ge65$ ) or gender.

Figure 3: Effect of Atorvastatin 80 mg/day vs. 10 mg/day on Time to Occurrence of Major Cardiovascular Events (TNT)



**TABLE 5. Overview of Efficacy Results in TNT** 

| Endpoint | 10 | astatin<br>mg<br>5006) | Atorvastatin<br>80 mg<br>(N=4995) | | HR* (95%CI) |
|---|---|---|---|---|---|
| PRIMARY ENDPOINT | n | (%) | n | (%) | |
| First major cardiovascular endpoint | 548 | (10.9) | 434 | (8.7) | 0.78 (0.69, 0.89) |
| Components of the Primary Endpoint | | | | | |
| CHD death | 127 | (2.5) | 101 | (2.0) | 0.80 (0.61, 1.03) |
| Non-fatal, non-procedure related MI | 308 | (6.2) | 243 | (4.9) | 0.78 (0.66, 0.93) |
| Resuscitated cardiac arrest | 26 | (0.5) | 25 | (0.5) | 0.96 (0.56, 1.67) |
| Stroke (fatal and non-fatal) | 155 | (3.1) | 117 | (2.3) | 0.75 (0.59, 0.96) |
| SECONDARY ENDPOINTS† | | | | | |
| First CHF with hospitalization | 164 | (3.3) | 122 | (2.4) | 0.74 (0.59, 0.94) |
| First PVD endpoint | 282 | (5.6) | 275 | (5.5) | 0.97 (0.83, 1.15) |
| First CABG or other coronary revascularization procedure <sup>‡</sup> | 904 | (18.1) | 667 | (13.4) | 0.72 (0.65, 0.80) |
| First documented angina endpoint <sup>‡</sup> | 615 | (12.3) | 545 | (10.9) | 0.88 (0.79, 0.99) |
| All-cause mortality | 282 | (5.6) | 284 | (5.7) | 1.01 (0.85, 1.19) |
| Components of All-Cause Mortality | | | | | |
| Cardiovascular death | 155 | (3.1) | 126 | (2.5) | 0.81 (0.64, 1.03) |
| Noncardiovascular death | 127 | (2.5) | 158 | (3.2) | 1.25 (0.99, 1.57) |
| Cancer death | 75 | (1.5) | 85 | (1.7) | 1.13 (0.83, 1.55) |
| Other non-CV death | 43 | (0.9) | 58 | (1.2) | 1.35 (0.91, 2.00) |
| Suicide, homicide, and other traumatic non-CV | | | | | |

Page 300 of 364

| death | 9 | (0.2) | 15 | (0.3) | 1.67 (0.73, 3.82) |
|-------|---|-------|----|-------|-------------------|
|-------|---|-------|----|-------|-------------------|

HR=hazard ratio; CHD=coronary heart disease; CI=confidence interval; MI=myocardial infarction; CHF=congestive heart failure; CV=cardiovascular; PVD=peripheral vascular disease; CABG=coronary artery bypass graft

Confidence intervals for the Secondary Endpoints were not adjusted for multiple comparisons

- \* Atorvastatin 80 mg: atorvastatin 10 mg
- † Secondary endpoints not included in primary endpoint
- Component of other secondary endpoints

Of the events that comprised the primary efficacy endpoint, treatment with atorvastatin calcium tablets 80 mg/day significantly reduced the rate of non-fatal, non-procedure related MI and fatal and non-fatal stroke, but not CHD death or resuscitated cardiac arrest (Table 5). Of the predefined secondary endpoints, treatment with atorvastatin calcium tablets 80 mg/day significantly reduced the rate of coronary revascularization, angina, and hospitalization for heart failure, but not peripheral vascular disease. The reduction in the rate of CHF with hospitalization was only observed in the 8% of patients with a prior history of CHF.

There was no significant difference between the treatment groups for all-cause mortality (Table 5). The proportions of subjects who experienced cardiovascular death, including the components of CHD death and fatal stroke, were numerically smaller in the atorvastatin calcium tablets 80 mg group than in the atorvastatin calcium tablets 10 mg treatment group. The proportions of subjects who experienced noncardiovascular death were numerically larger in the atorvastatin calcium tablets 80 mg group than in the atorvastatin calcium tablets 10 mg treatment group.

In the Incremental Decrease in Endpoints Through Aggressive Lipid Lowering Study (IDEAL), treatment with atorvastatin calcium tablets 80 mg/day was compared to treatment with simvastatin 20–40 mg/day in 8,888 subjects up to 80 years of age with a history of CHD to assess whether reduction in CV risk could be achieved. Patients were mainly male (81%), white (99%) with an average age of 61.7 years, and an average LDL-C of 121.5 mg/dL at randomization; 76% were on statin therapy. In this prospective, randomized, open-label, blinded endpoint (PROBE) trial with no run-in period, subjects were followed for a median duration of 4.8 years. The mean LDL-C, TC, TG, HDL, and non-HDL cholesterol levels at Week 12 were 78, 145, 115, 45, and 100 mg/dL during treatment with 80 mg of atorvastatin calcium tablets and 105, 179, 142, 47, and 132 mg/dL during treatment with 20–40 mg of simvastatin

There was no significant difference between the treatment groups for the primary endpoint, the rate of first major coronary event (fatal CHD, non-fatal MI, and resuscitated cardiac arrest): 411 (9.3%) in the atorvastatin calcium tablets 80 mg/day group vs. 463 (10.4%) in the simvastatin 20–40 mg/day group, HR 0.89, 95% CI (0.78, 1.01), p=0.07.

There were no significant differences between the treatment groups for all-cause mortality: 366 (8.2%) in the atorvastatin calcium tablets 80 mg/day group vs. 374 (8.4%) in the simvastatin 20–40 mg/day group. The proportions of subjects who experienced CV or non-CV death were similar for the atorvastatin calcium tablets 80 mg group and the simvastatin 20–40 mg group.

# 14.2 Hyperlipidemia (Heterozygous Familial and Nonfamilial) and Mixed Dyslipidemia (*Fredrickson* Types IIa and IIb)

Atorvastatin reduces total-C, LDL-C, VLDL-C, apo B, and TG, and increases HDL-C in patients with hyperlipidemia and mixed dyslipidemia. Therapeutic response is seen within 2 weeks, and maximum response is usually achieved within 4 weeks and maintained during chronic therapy.

Atorvastatin calcium tablets are effective in a wide variety of patient populations with hyperlipidemia, with and without hypertriglyceridemia, in men and women, and in the elderly.

In two multicenter, placebo-controlled, dose-response studies in patients with hyperlipidemia, atorvastatin calcium tablets given as a single dose over 6 weeks, significantly reduced total-C, LDL-C, apo B, and TG. (Pooled results are provided in Table 6.)

TABLE 6. Dose Response in Patients With Primary Hyperlipidemia (Adjusted Mean % Change From Baseline)\*

| Dose | N | TC | LDL-C | Apo B | TG | HDL-C | Non-HDL-<br>C/ HDL-C |
|---------|----|-----|-------|-------|-----|-------|----------------------|
| Placebo | 21 | 4 | 4 | 3 | 10 | -3 | 7 |
| 10 | 22 | -29 | -39 | -32 | -19 | 6 | -34 |
| 20 | 20 | -33 | -43 | -35 | -26 | 9 | -41 |
| 40 | 21 | -37 | -50 | -42 | -29 | 6 | -45 |
| 80 | 23 | -45 | -60 | -50 | -37 | 5 | -53 |

<sup>\*</sup> Results are pooled from 2 dose-response studies.

In patients with *Fredrickson* Types IIa and IIb hyperlipoproteinemia pooled from 24 controlled trials, the median (25<sup>th</sup> and 75<sup>th</sup> percentile) percent changes from baseline in HDL-C for atorvastatin calcium tablets 10, 20, 40, and 80 mg were 6.4 (-1.4, 14), 8.7 (0, 17), 7.8 (0, 16), and 5.1 (-2.7, 15), respectively. Additionally, analysis of the pooled data demonstrated consistent and significant decreases in total-C, LDL-C, TG, total-C/HDL-C, and LDL-C/HDL-C.

In three multicenter, double-blind studies in patients with hyperlipidemia, atorvastatin was compared to other statins. After randomization, patients were treated for 16 weeks with either atorvastatin calcium tablets 10 mg per day or a fixed dose of the comparative agent (Table 7).

TABLE 7. Mean Percentage Change From Baseline at Endpoint (Double-Blind, Randomized, Active-Controlled Trials)

| | | | Controlled | 1 1 1 a 1 5 <i>j</i> | | | |
|---|---|---|---|---|---|---|---|
| Treatment (Daily Dose) | N | Total-C | LDL-C | Apo B | TG | HDL-C | Non-HDL-<br>C/ HDL-C |
| Study 1 | | | | | | | |
| Atorvastatin 10 mg | 707 | -27* | -36* | -28* | -17* | +7 | -37* |
| Lovastatin 20 mg | 191 | -19 | -27 | -20 | -6 | +7 | -28 |
| 95% CI for Diff <sup>†</sup> | | -9.2, -6.5 | -10.7, -7.1 | -10.0, -6.5 | -15.2, -7.1 | -1.7, 2.0 | -11.1, -7.1 |
| Study 2 | | | | | | | |
| Atorvastatin 10 mg | 222 | -25‡ | -35‡ | -27‡ | -17‡ | +6 | -36‡ |
| Pravastatin 20 mg | 77 | -17 | -23 | -17 | -9 | +8 | -28 |
| 95% CI for Diff <sup>†</sup> | | -10.8, -6.1 | -14.5, -8.2 | -13.4, -7.4 | -14.1, -0.7 | -4.9, 1.6 | -11.5, -4.1 |
| Study 3 | | | | | | | |
| Atorvastatin 10 mg | 132 | -29§ | -37§ | -34§ | -23§ | +7 | -39§ |
| Simvastatin 10 mg | 45 | -24 | -30 | -30 | -15 | +7 | -33 |
| 95% CI for Diff <sup>†</sup> | | -8.7, -2.7 | -10.1, -2.6 | -8.0, -1.1 | -15.1, -0.7 | -4.3, 3.9 | -9.6, -1.9 |

<sup>\*</sup> Significantly different from lovastatin, ANCOVA,  $p \le 0.05$ 

The impact on clinical outcomes of the differences in lipid-altering effects between treatments shown in Table 7 is

<sup>†</sup> A negative value for the 95% CI for the difference between treatments favors atorvastatin for all except HDL-C, for which a positive value favors atorvastatin. If the range does not include 0, this indicates a statistically significant difference.

 $<sup>\</sup>ddagger$  Significantly different from pravastatin, ANCOVA, p  $\leq$  0.05

<sup>§</sup> Significantly different from simvastatin, ANCOVA, p ≤0.05

not known. Table 7 does not contain data comparing the effects of atorvastatin 10 mg and higher doses of lovastatin, pravastatin, and simvastatin. The drugs compared in the studies summarized in the table are not necessarily interchangeable.

# 14.3 Hypertriglyceridemia (Fredrickson Type IV)

The response to atorvastatin in 64 patients with isolated hypertriglyceridemia treated across several clinical trials is shown in the table below (Table 8). For the atorvastatin calcium tablets-treated patients, median (min, max) baseline TG level was 565 (267–1502).

TABLE 8. Combined Patients With Isolated Elevated TG: Median (min, max) Percentage Change From Baseline

| | | ***** | | |
|---|---|---|---|---|
| | Placebo<br>(N=12) | atorvastatin 10 mg<br>(N=37) | atorvastatin 20 mg<br>(N=13) | atorvastatin 80 mg<br>(N=14) |
| Triglycerides | -12.4 (-36.6, 82.7) | -41.0 (-76.2, 49.4) | -38.7 (-62.7, 29.5) | -51.8 (-82.8, 41.3) |
| Total-C | -2.3 (-15.5, 24.4) | -28.2 (-44.9, -6.8) | -34.9 (-49.6, -15.2) | -44.4 (-63.5, -3.8) |
| LDL-C | 3.6 (-31.3, 31.6) | -26.5 (-57.7, 9.8) | -30.4 (-53.9, 0.3) | -40.5 (-60.6, -13.8) |
| HDL-C | 3.8 (-18.6, 13.4) | 13.8 (-9.7, 61.5) | 11.0 (-3.2, 25.2) | 7.5 (-10.8, 37.2) |
| VLDL-C | -1.0 (-31.9, 53.2) | -48.8 (-85.8, 57.3) | -44.6 (-62.2, -10.8) | -62.0 (-88.2, 37.6) |
| non-HDL-C | -2.8 (-17.6, 30.0) | -33.0 (-52.1, -13.3) | -42.7 (-53.7, -17.4) | -51.5 (-72.9, -4.3) |

# 14.4 Dysbetalipoproteinemia (Fredrickson Type III)

The results of an open-label crossover study of 16 patients (genotypes: 14 apo E2/E2 and 2 apo E3/E2) with dysbetalipoproteinemia (*Fredrickson* Type III) are shown in the table below (Table 9).

TABLE 9. Open-Label Crossover Study of 16 Patients With Dysbetalipoproteinemia (Fredrickson Type III)

| | | Median % Change (min, max) | |
|---|---|---|---|
| | Median (min, max) at<br>Baseline (mg/dL) | atorvastatin 10<br>mg | atorvastatin 80<br>mg |
| Total-C | 442 (225, 1320) | -37 (-85, 17) | -58 (-90, -31) |
| Triglycerides | 678 (273, 5990) | -39 (-92, -8) | -53 (-95, -30) |
| IDL-C + VLDL-C | 215 (111, 613) | -32 (-76, 9) | -63 (-90, -8) |
| non-HDL-C | 411 (218, 1272) | -43 (-87, -19) | -64 (-92, -36) |

# 14.5 Homozygous Familial Hypercholesterolemia

In a study without a concurrent control group, 29 patients ages 6 to 37 years with homozygous FH received maximum daily doses of 20 to 80 mg of atorvastatin calcium tablets. The mean LDL-C reduction in this study was 18%. Twenty-five patients with a reduction in LDL-C had a mean response of 20% (range of 7% to 53%, median of 24%); the remaining 4 patients had 7% to 24% increases in LDL-C. Five of the 29 patients had absent LDL-receptor function. Of these, 2 patients also had a portacaval shunt and had no significant reduction in LDL-C. The remaining 3 receptor-negative patients had a mean LDL-C reduction of 22%.

# 14.6 Heterozygous Familial Hypercholesterolemia in Pediatric Patients

In a double-blind, placebo-controlled study followed by an open-label phase, 187 boys and postmenarchal girls 10–17 years of age (mean age 14.1 years) with heterozygous familial hypercholesterolemia (FH) or severe hypercholesterolemia, were randomized to atorvastatin calcium tablets (n=140) or placebo (n=47) for 26 weeks and then all received atorvastatin calcium tablets for 26 weeks. Inclusion in the study required 1) a baseline LDL-C level ≥ 190 mg/dL or 2) a baseline LDL-C level ≥ 160 mg/dL and positive family history of FH or documented premature cardiovascular disease in a first or second-degree relative. The mean baseline LDL-C value was 218.6 mg/dL (range: 138.5–385.0 mg/dL) in the atorvastatin calcium tablets group compared to 230.0 mg/dL (range: 160.0–324.5 mg/dL) in the placebo group. The dosage of atorvastatin calcium tablets (once daily) was 10 mg for the first 4 weeks and uptitrated to 20 mg if the LDL-C level was > 130 mg/dL. The number of atorvastatin calcium tablets-treated patients who required uptitration to 20 mg after Week 4 during the double-blind phase was 78 (55.7%).

Atorvastatin significantly decreased plasma levels of total-C, LDL-C, triglycerides, and apolipoprotein B during the 26-week double-blind phase (see Table 10).

TABLE 10. Lipid-altering Effects of Atorvastatin in Adolescent Boys and Girls with Heterozygous Familial Hypercholesterolemia or Severe Hypercholesterolemia (Mean Percentage Change From Baseline at Endpoint in Intention-to-Treat Population)

| DOSAGE | N | Total-C | LDL-C | HDL-C | TG | Apolipoprotein<br>B |
|--------------|-----|---------|-------|-------|-------|---------------------|
| Placebo | 47 | -1.5 | -0.4 | -1.9 | 1.0 | 0.7 |
| Atorvastatin | 140 | -31.4 | -39.6 | 2.8 | -12.0 | -34.0 |

The mean achieved LDL-C value was 130.7 mg/dL (range: 70.0–242.0 mg/dL) in the atorvastatin group compared to 228.5 mg/dL (range: 152.0–385.0 mg/dL) in the placebo group during the 26-week double-blind phase.

The safety and efficacy of doses above 20 mg have not been studied in controlled trials in children. The long-term efficacy of atorvastatin therapy in childhood to reduce morbidity and mortality in adulthood has not been established.

### 15 REFERENCES

<sup>1</sup>National Cholesterol Education Program (NCEP): Highlights of the Report of the Expert Panel on Blood Cholesterol Levels in Children and Adolescents, *Pediatrics*. 89(3):495–501. 1992.

### 16 HOW SUPPLIED/STORAGE AND HANDLING

10 mg tablets: coded "PD 155" on one side and "10" on the other.

NDC 59762-0155-1 bottles of 90 NDC 59762-0155-2 bottles of 1000

20 mg tablets: coded "PD 156" on one side and "20" on the other.

NDC 59762-0156-1 bottles of 90 NDC 59762-0156-2 bottles of 1000

40 mg tablets: coded "PD 157" on one side and "40" on the other.

NDC 59762-0157-1 bottles of 90

NDC 59762-0157-2 bottles of 500

80 mg tablets: coded "PD 158" on one side and "80" on the other.

NDC 59762-0158-1 bottles of 90 NDC 59762-0158-2 bottles of 500

### **Storage**

Store at controlled room temperature  $20 - 25^{\circ}\text{C}$  (68 - 77°F) [see USP].

# 17 PATIENT COUNSELING INFORMATION

Patients taking atorvastatin calcium tablets should be advised that cholesterol is a chronic condition and they should adhere to their medication along with their National Cholesterol Education Program (NCEP)-recommended diet, a regular exercise program as appropriate, and periodic testing of a fasting lipid panel to determine goal attainment.

Patients should be advised about substances they should not take concomitantly with atorvastatin [see Warnings and Precautions (5.1)]. Patients should also be advised to inform other healthcare professionals prescribing a new medication that they are taking atorvastatin calcium tablets.

### 17.1 Muscle Pain

All patients starting therapy with atorvastatin calcium tablets should be advised of the risk of myopathy and told to report promptly any unexplained muscle pain, tenderness, or weakness particularly if accompanied by malaise or fever or if these muscle signs or symptoms persist after discontinuing atorvastatin calcium tablets. The risk of this occurring is increased when taking certain types of medication or consuming larger quantities (>1 liter) of grapefruit juice. They should discuss all medication, both prescription and over the counter, with their healthcare professional.

# 17.2 Liver Enzymes

It is recommended that liver enzyme tests be performed before the initiation of atorvastatin calcium tablets and if signs or symptoms of liver injury occur. All patients treated with atorvastatin calcium tablets should be advised to report promptly any symptoms that may indicate liver injury, including fatigue, anorexia, right upper abdominal discomfort, dark urine, or jaundice.

### 17.3 Pregnancy

Women of childbearing age should be advised to use an effective method of birth control to prevent pregnancy while using atorvastatin calcium tablets. Discuss future pregnancy plans with your patients, and discuss when to stop atorvastatin calcium tablets if they are trying to conceive. Patients should be advised that if they become pregnant, they should stop taking atorvastatin calcium tablets and call their healthcare professional.

# 17.4 Breast-feeding

Women who are breastfeeding should be advised to not use atorvastatin calcium tablets. Patients who have a lipid disorder and are breast-feeding, should be advised to discuss the options with their healthcare professional.



LAB-0644-3.0

### PATIENT INFORMATION

### **Atorvastatin Calcium Tablets**

Read the Patient Information that comes with atorvastatin calcium tablets before you start taking it and each time you get a refill. There may be new information. This leaflet does not take the place of talking with your doctor about your condition or treatment.

If you have any questions about atorvastatin calcium tablets, ask your doctor or pharmacist.

### What Are Atorvastatin Calcium Tablets?

Atorvastatin calcium is a prescription medicine that lowers cholesterol in your blood. It lowers the LDL-C ("bad" cholesterol) and triglycerides in your blood. It can raise your HDL-C ("good" cholesterol) as well. Atorvastatin calcium tablets are for adults and children over 10 whose cholesterol does not come down enough with exercise and a low-fat diet alone.

Atorvastatin calcium tablets can lower the risk for heart attack, stroke, certain types of heart surgery, and chest pain in patients who have heart disease or risk factors for heart disease such as:

• age, smoking, high blood pressure, low HDL-C, heart disease in the family.

Atorvastatin calcium tablets can lower the risk for heart attack or stroke in patients with diabetes and risk factors such as:

• eye problems, kidney problems, smoking, or high blood pressure.

Atorvastatin calcium tablets start to work in about 2 weeks.

### What is Cholesterol?

Cholesterol and triglycerides are fats that are made in your body. They are also found in foods. You need some cholesterol for good health, but too much is not good for you. Cholesterol and triglycerides can clog your blood vessels. It is especially important to lower your cholesterol if you have heart disease, smoke, have diabetes or high blood pressure, are older, or if heart disease starts early in your family.

### Who Should Not Take Atorvastatin Calcium Tablets?

Do not take atorvastatin calcium tablets if you:

- are pregnant or think you may be pregnant, or are planning to become pregnant. Atorvastatin calcium tablets may harm your unborn baby. If you get pregnant, stop taking atorvastatin calcium tablets and call your doctor right away.
- are breast feeding. Atorvastatin calcium tablets can pass into your breast milk and may harm your baby.
- have liver problems.
- are allergic to atorvastatin calcium tablets or any of its ingredients. The active ingredient is atorvastatin. See the end of this leaflet for a complete list of ingredients in atorvastatin calcium tablets.

Atorvastatin calcium tablets have not been studied in children under 10 years of age.

### **Before You Start Atorvastatin Calcium Tablets**

Tell your doctor if you:

have muscle aches or weakness

drink more than 2 glasses of alcohol daily

- have diabetes
- have a thyroid problem
- have kidney problems

Some medicines should not be taken with atorvastatin calcium tablets. Tell your doctor about all the medicines you take, including prescription and non-prescription medicines, vitamins, and herbal supplements. Atorvastatin calcium tablets and certain other medicines can interact causing serious side effects. Especially tell your doctor if you take medicines for:

- your immune system
- cholesterol
- infections
- birth control
- heart failure
- HIV or AIDS

Know all the medicines you take. Keep a list of them with you to show your doctor and pharmacist.

### **How Should I Take Atorvastatin Calcium Tablets?**

- Take atorvastatin calcium tablets exactly as prescribed by your doctor. Do not change your dose or stop atorvastatin calcium tablets without talking to your doctor. Your doctor may do blood tests to check your cholesterol levels during your treatment with atorvastatin calcium tablets. Your dose of atorvastatin calcium tablets may be changed based on these blood test results.
- Take atorvastatin calcium tablets each day at any time of day at about the same time each day. Atorvastatin calcium tablets can be taken with or without food.
  - Don't break atorvastatin calcium tablets before taking.
- Your doctor should start you on a low-fat diet before giving you atorvastatin calcium tablets. Stay on this low-fat diet when you take atorvastatin calcium tablets.
- If you miss a dose of atorvastatin calcium tablets, take it as soon as you remember. Do not take atorvastatin calcium tablets if it has been more than 12 hours since you missed your last dose. Wait and take the next dose at your regular time. Do not take 2 doses of atorvastatin calcium tablets at the same time.
- If you take too much atorvastatin calcium tablets or overdose, call your doctor or Poison Control Center right away. Or go to the nearest emergency room.

# What Should I Avoid While Taking Atorvastatin Calcium Tablets?

- Talk to your doctor before you start any new medicines. This includes prescription and non-prescription medicines, vitamins, and herbal supplements. Atorvastatin calcium tablets and certain other medicines can interact causing serious side effects.
- Do not get pregnant. If you get pregnant, stop taking atorvastatin calcium tablets right away and call your doctor.

# What are the Possible Side Effects of Atorvastatin Calcium Tablets?

Atorvastatin calcium tablets can cause serious side effects. These side effects have happened only to a small number of people. Your doctor can monitor you for them. These side effects usually go away if your dose is lowered or atorvastatin calcium tablets are stopped.

### These serious side effects include:

- **Muscle problems.** Atorvastatin calcium tablets can cause serious muscle problems that can lead to kidney problems, including kidney failure. You have a higher chance for muscle problems if you are taking certain other medicines with atorvastatin calcium tablets.
- **Liver problems.** Your doctor should do blood tests to check your liver before you start taking atorvastatin calcium tablets, and if you have symptoms of liver problems while you take atorvastatin calcium tablets. Call your doctor right away if you have the following symptoms of liver problems:
  - feel tired or weak
  - loss of appetite

- upper belly pain
- dark amber colored urine
- yellowing of your skin or the whites of your eyes

# Call your doctor right away if you have:

- muscle problems like weakness, tenderness, or pain that happen without a good reason, especially if you also have a fever or feel more tired than usual. This may be an early sign of a rare muscle problem.
- muscle problems that do not go away even after your doctor has advised you to stop taking atorvastatin calcium tablets. Your doctor may do further tests to diagnose the cause of your muscle problems.
- allergic reactions including swelling of the face, lips, tongue, and/or throat that may cause difficulty in breathing or swallowing which may require treatment right away.
- nausea and vomiting.
- passing brown or dark-colored urine.
- you feel more tired than usual
- your skin and whites of your eyes get yellow.
- stomach pain.
- allergic skin reactions.

In clinical studies, patients reported the following common side effects while taking atorvastatin calcium tablets: diarrhea, upset stomach, muscle and joint pain, and alterations in some laboratory blood tests.

The following additional side effects have been reported with atorvastatin calcium tablets: tiredness, tendon problems, memory loss, and confusion.

Talk to your doctor or pharmacist if you have side effects that bother you or that will not go away.

These are not all the side effects of atorvastatin calcium tablets. Ask your doctor or pharmacist for a complete list.

### How do I store Atorvastatin Calcium Tablets?

- Store atorvastatin calcium tablets at room temperature, 68 to 77°F (20 to 25°C).
- Do not keep medicine that is out of date or that you no longer need.
- Keep atorvastatin calcium tablets and all medicines out of the reach of children. Be sure that if you throw medicine away, it is out of the reach of children.

### **General Information about Atorvastatin Calcium Tablets**

Medicines are sometimes prescribed for conditions that are not mentioned in patient information leaflets. Do not use atorvastatin calcium tablets for a condition for which it was not prescribed. Do not give atorvastatin calcium tablets to other people, even if they have the same problem you have. It may harm them.

This leaflet summarizes the most important information about atorvastatin calcium tablets. If you would like more information, talk with your doctor. You can ask your doctor or pharmacist for information about atorvastatin calcium tablets that is written for health professionals.

# What are the Ingredients in Atorvastatin Calcium Tablets?

**Active Ingredient:** atorvastatin calcium

**Inactive Ingredients:** calcium carbonate, USP; candelilla wax, FCC; croscarmellose sodium, NF; hydroxypropyl cellulose, NF; lactose monohydrate, NF; magnesium stearate, NF; microcrystalline cellulose, NF; Opadry White YS-1-7040 (hypromellose, polyethylene glycol, talc, titanium dioxide); polysorbate 80, NF; simethicone emulsion.



Revised: 3/2015 Greenstone LLC

# APPENDIX F. 747-209 PROTOCOL VERSION 2 SUMMARY OF CHANGES

# **Background**

Protocol 747-209 has been prepared as a Phase 2 trial to evaluate the effect of OCA on LDL metabolism in subjects with biopsy-confirmed NASH and to assess the ability of atorvastatin to modulate this effect.

Protocol 747-209 Version 2 (dated 22 October 2015) incorporates suggestions made by the FDA regarding the 747-303 protocol that are also relevant to this study.

### Rationale

Protocol 747-209 Version 2 has been prepared to:

- 1. Clarify stopping rules for subjects presenting with a CTCAE of ≥Grade 3, per FDA's comments on the 747-303 protocol.
- 2. Clarify that subjects discontinued due to significant drug-induced liver injury will be followed until the AE has resolved, stabilized, or is not of clinical concern.
- 3. Clarify atorvastatin safety profile.
- 4. Include a description for the cardiovascular events adjudication committee, and add Appendix D to define major cardiovascular events.

In addition, Protocol 747-209 Version 2 also:

- 1. Clarifies contraception requirements.
- 2. Adds additional exploratory objectives: markers of cardiovascular safety
- 3. Clarifies exclusion criteria related to chronic liver diseases at Screening.
- 4. Removes the requirement that a study site must have prior experience treating patients with NASH to participate in this study.
- 5. Clarifies PD assessments; markers of inflammation, fibrosis, and apoptosis; and PK assessments in the Schedule of Study Procedures tables, and in the text.
- 6. Clarifies timepoints for PK blood sample collection.
- 7. Corrects the title of Appendix A to reflect ACA/AHA guidance for the use of statins.

# **Summary of Changes**

The following revisions were made to the protocol in Protocol Version 2.

Note: (1) Revised text in Version 2 is indicated in bold font, and the text deleted from the Original protocol is crossed out in the table below. (2) Minor/editorial changes, including additional abbreviations defined are not listed individually in the summary table below.

| Section | Original Text (Original protocol) | | | Revised Text (Version 2) |
|---|---|---|---|---|
| Global changes<br>(throughout<br>document) | | | CK-18-M65 added in addition to CK-18-M30 assessme<br>marker for hepatic apoptosis and fibrosis under Explor<br>Endpoints | |
| | | | | ty Monitoring Committee (DSMC) changed to ing Committee (DMC) |
| Study Personnel | Emergency Co | ntact Information | Medical Monit | tor |
| Contact<br>Information<br>(Cover Page) | Medical Monitor — 24-hour Emergency Reporting | | Investigators are encouraged to call the NASH medical monitor hotline at +1 844 250 6396 or send an email to t NASH medical monitor at NASH209@interceptpharma.com with safety questions these lines of contact are monitored 24 hours a day. | |
| | Contact: | Roya Hooshmand-Rad, MD PhD,<br>Executive Director, Clinical Research<br>Intercept Pharmaceuticals, Inc.<br>(Intercept) | Primary<br>Medical<br>Monitor<br>Contact: | Roya Hooshmand-Rad, MD PhD<br>Executive Director, Clinical Research<br>Intercept Pharmaceuticals, Inc. (Intercept |
| | Telephone: | <del>+1 844 250 6396</del> | Email: | rhooshmand-rad@interceptpharma.com |
| | Email: | rhooshmand-<br>rad@interceptpharma.com | | |
| | SAE Fax: | <del>+ 1 800 497 8521</del> | | |
| | SAE Email: | sae@interceptpharma.com | | |
| | Or if Not Avai | <del>lable:</del> | | |

| Section | Original | Text (Original protocol) | Rev | Revised Text (Version 2) |
|---|---|---|---|---|
| | Med Inte Telephone: +1: | bara Scholz, MD, dical Director, Drug Safety rcept 844 250 6396 para.scholz@interceptpharma.com | Secondary Contact: Telephone: Email: | Barbara Scholz, MD, Medical Director, Drug Safety Intercept +1 858 353 1350 (Pacific time zone) barbara.scholz@interceptpharma.co m |
| Synopsis<br>(Exploratory<br>Objectives) | Liver<br>biochemistry and<br>markers of liver<br>function | Albumin, ALP, ALT, AST, , direct bilirubin, GGT, INR, total bilirubin | ` ` | Albumin, ALP (isoenzymes), ALT, AST, , direct bilirubin, GGT, INR, total bilirubin (me) was also added to the list of ts in Section 11.1 (Table 4) and 9). |
| Synopsis (Exploratory Objectives) And Section 6.3 (Exploratory Objectives) | | | Cardiovascular risk<br>[FRS] and Reynolds | scores (eg, Framingham Risk Score<br>score) |
| Synopsis (Methodology) <u>And</u> Section 7.1 Overall Study Design (Double-Blind Phase) | | | atorvastatin during a expected to attend so followed through the Subjects who discomblind phase are eligit double-blind phase a discretion of the Investment | tinue investigational product or<br>the double-blind phase are still<br>cheduled study visits and are to be<br>e Week 16 Visit.<br>tinue atorvastatin during the double-<br>ble to continue OCA during the<br>and enroll into the LTSE at the<br>estigator, provided they continue to<br>ria #4 (LDL <200 mg/dL). |

|---|---|---|
| Synopsis (Study Design Diagram) And Section 7.1.1 Study Design, Figure 1 | | Footnote Added: \$\Delta\$ = Telephone safety contact at Week 6, Week 10, and Week 14 |
| Synopsis (Key Inclusion Criteria) And Section 8.2 Subject Inclusion Criteria | <ul> <li>6. Contraception: Female subjects of childbearing potential must use ≥1 effective method of contraception during both the double-blind and LTSE phases of the study and 4 weeks following the last dose of investigational product or at study termination (whichever is greater). Effective methods of contraception are considered to be those listed as follows:</li> <li>Double-barrier method, ie, (a) condom (male or female) or (b) diaphragm, with spermicide; or</li> <li>Intrauterine device; or</li> <li>Vasectomy (partner); or</li> <li>Hormonal (eg, contraceptive pill, patch, intramuscular implant or injection); or</li> <li>Abstinence, if in line with the preferred and usual lifestyle of the subject</li> </ul> | <ul> <li>6. Contraception: Female subjects of childbearing potential must use ≥1 effective method of contraception during the study and until 30 days following the last dose of investigational product. Effective methods of contraception are considered to be those listed below.</li> <li>Double-barrier method, ie, (a) condom (male or female) or (b) diaphragm, with spermicide</li> <li>Intrauterine device</li> <li>Vasectomy (partner)</li> <li>Hormonal (eg, contraceptive pill, patch, intramuscular implant or injection)</li> <li>Abstinence (defined as refraining from heterosexual intercourse)</li> </ul> |
| Synopsis<br>(Key Exclusion<br>Criteria) | 3.LDL cholesterol ≥190 mg/dL and already on statin therapy at Screening Visit 1. | 3.LDL cholesterol ≥190 mg/dL and already on statin therapy at Screening Visit 1. |
| And Section 8.3 Subject Exclusion Criteria | <ul> <li>10. Evidence of other forms of chronic liver disease including but not limited to:</li> <li>Concomitant hepatitis B or C virus infection</li> <li>•</li> </ul> | <ul> <li>10. Evidence of other forms of chronic liver disease including but not limited to:</li> <li>Positive test result at Screening for hepatitis B surface antigen or hepatitis C antibody (and positive hepatitis C virus [HCV] ribonucleic acid [RNA])</li> </ul> |

|---|---|
| 11. Presence of clinically significant hepatic decompensation, including: •History of liver transplant, current placement on a liver transplant list, or current Model for End-Stage Liver Disease (MELD) score >12. Subjects who are placed on a transplant list despite a relatively early disease stage (eg, per regional guidelines) may be eligible as long as they do not meet any of the other exclusion criteria. •History (within the past 12 months) or presence of: oVariceal bleed oUncontrolled ascites oHepatic encephalopathy oSpontaneous bacterial peritonitis oHepatorenal or hepatopulmonary syndromes | 11. History of liver transplant, current placement on a liver transplant list, or current Model for End-Stage Liver Disease (MELD) score >12. Subjects who are placed on a transplant list despite a relatively early disease stage (eg, per regional guidelines) may be eligible as long as they do not meet any of the other exclusion criteria. |
| | 12. Presence of hepatic decompensation, including: - Gastroesophageal varices - Ascites - Hepatic encephalopathy - Spontaneous bacterial peritonitis - Hepatorenal or hepatopulmonary syndromes |
| 14. Creatine phosphokinase >5x ULN at any Screening visit. | 14. Creatine phosphokinase >5x ULN at Screening Visit 2. |
| 19a. Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) | 19a. <b>Peripheral or</b> Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) |
| | Note: Exclusion criteria numbered 12 through 27 in the Original Protocol updated to numbers 13 through 28 in Version 2 as a result of new exclusion criteria number 12 above. |

| Section | Original | Text (Original protocol) | I | Revised Text (Version 2) |
|---|---|---|---|---|
| Synopsis | Secondary Endpoints | | Secondary Endpoin | nts |
| (Statistical Methods) | Safety and tolerability | TEAEs, physical exams, ECGs, vital signs, clinical laboratory assessments (including lipid profile changes) | Safety and tolerability | TEAEs (including cardiovascular events), physical exams, ECGs, vital signs, clinical laboratory assessments (including lipid profile changes) |
| Synopsis | Exploratory Endpoint | S | Exploratory Endpo | ints |
| (Statistical Methods) And | Liver biochemistry<br>and markers of<br>liver function | Albumin, ALP, ALT, AST, ereatinine, GGT, total bilirubin, eonjugated (direct)-bilirubin, INR | Liver biochemistr<br>and markers of liv<br>function | |
| Section 11.1<br>Efficacy<br>Assessments<br>(Table 4) | Marker for hepatic apoptosis and fibrosis | CK-18-M30 | Marker for hepati<br>apoptosis and<br>fibrosis | c CK-18-M30 and CK-18-M65 |
| | | | Cardiovascular risk scores | FRS and Reynolds scores |
| Synopsis (Sample Size Justification) And Section 13.2 Determination of Sample Size | It is the intent of this study to characterize the components of LDL metabolism (cholesterol concentration, particle size, particle concentration) in subjects with NASH before and after treatment with OCA and to assess the changes induced by HMG Coenzyme A reductase inhibitor (atorvastatin) therapy. Assuming a 22 U/L increase from baseline with a standard deviation of 20 in LDL in the OCA 25 mg group, a sample size of 20 subjects per group will provide greater than 99.9% power to demonstrate the statistically significant difference of LDL increase from baseline with a 2-sided type I error of 0.05 | | LDL metabolism (a particle concentration after treatment with by HMG Coenzym therapy. Assuming standard deviation without atorvasta based on data from group will provide the statistically significant concentration. | cholesterol concentration, particle size, ion) in subjects with NASH before and in OCA and to assess the changes induced as A reductase inhibitor (atorvastatin) g, 22 mg/dL increase from baseline with a of 24 in LDL in the OCA 25 mg group tin therapy after 16 weeks of treatment in FLINT, a sample size of 20 subjects per greater than 97.3% power to demonstrate inificant difference of LDL increase from ided type I error of 0.05. |
| Section 5.6.4.1<br>Rationale for | cardiovascular disease | de subjects with existing<br>e (including but not limited to stable<br>evious myocardial infarction or | disease (including | clude subjects with existing cardiovascular<br>but not limited to stable or unstable angina,<br>al infarction or stroke or a previous |


|---|---|---|
| statin withdrawal<br>(Paragraph 5) | stroke or a previous coronary revascularization procedure), significant dyslipidemia (as defined by LDL >190 mg/dL) despite the use of statin therapy, unstable hypertension, and familial hypercholesterolemia. | <b>peripheral or</b> coronary revascularization procedure), significant dyslipidemia (as defined by LDL ≥190 mg/dL) despite the use of statin therapy, unstable hypertension, and familial hypercholesterolemia |
| Section 5.8.<br>Summary of<br>Known Potential<br>Risks with<br>Atorvastatin | (Section 5.8 added to Version 2) | Muscle complaints are the most frequent adverse reports among patients treated with statins, with the most severe side effects including myopathy and rhabdomyolysis. The Statin Muscle Safety Task Force (Rosenson 2014) has provided a classification of the spectrum of statin-associated muscle AEs that may be seen in clinical practice and can be used in characterizing reports of muscle-related events. |
| | | a. Myalgia – unexplained muscle discomfort often described as "flu-like" symptoms |
| | | <ul> <li>Muscle aches</li> </ul> |
| | | <ul> <li>Muscle soreness</li> </ul> |
| | | <ul> <li>Muscle stiffness</li> </ul> |
| | | <ul> <li>Muscle tenderness</li> </ul> |
| | | <ul> <li>Muscle cramps with or shortly after exercise (not nocturnal cramping)</li> </ul> |
| | | b. Myopathy – muscle weakness (not attributed to pain and not necessarily associated with elevated CPK) |
| | | c. Myositis – muscle inflammation |
| | | d. Myonecrosis – muscle enzyme elevations or hyperCPKemia |
| | | <ul> <li>Mild &gt;3x baseline or ULN</li> </ul> |
| | | <ul> <li>Moderate ≥10x baseline or ULN</li> </ul> |
| | | <ul> <li>Severe ≥50x baseline or ULN</li> </ul> |

|---|
| e. Clinical Rhabdomyolysis - Myonecrosis with myoglobinuria or acute renal failure (increase in serum creatinine ≥0.5 mg/dL |
| There is no evidence that these muscle-related AEs are a continuum beginning with myalgia and progressing to more severe manifestations of myopathy; rather events occur independent of each other. Myalgia events, with frequencies ranging from 1% to 5% in clinical trials to 11% to 29% in observational cohorts, typically occur within 1 month of statin initiation and resolve within 2 weeks of statin cessation (Rosenson 2014). Retrospective analyses have suggested that patients who discontinue statins due to intolerance are able to tolerate statins long-term following re-challenge (Zhang 2013, Mampuya 2013). |
| Historically, statins have been associated with biochemical abnormalities of liver function, but available data suggest that increases in liver transaminases associated with statins are asymptomatic and generally reversible (Desai 2014). In the absence of liver disease, US guidelines (Stone 2013) recommend that baseline transaminase levels should be checked before initiating statin therapy and subsequent testing should only be done in the presence of symptoms suggestive of hepatic disease. As this study is being conducted in subjects with confirmed NASH, liver enzymes will be frequently monitored and Section 8.4.1.2, Section 8.4.1.3, and Appendix B provide detailed guidance for handling elevated liver biochemistry values. |
| Statins modestly increase the risk of type 2 diabetes mellitus in individuals with risk factors for diabetes. Individuals receiving statin therapy should be evaluated for new-onset diabetes according to the current diabetes screening guidelines (American Diabetes Association 2013). |

|---|---|---|
| | | Confusion and memory loss have been reported with statins, but medical evidence supporting a causal effect is weak or nonexistent (Simic 2015). However, any reports of cognitive events should be appropriately evaluated, particularly in individuals whose symptoms persist despite statin discontinuation. In this study, any AEs (including signs and symptoms described above) regardless of relationship to investigational product or study medication, must be documented appropriately (See Section 12) |
| 7.1<br>Overall Study<br>Design<br>(Table 1) | | Added Week 6 (Contact), Week 10 (Contact), and Week 14 (Contact) with associated X in AEs, Prior and Concomitant Medications, and Collect bottles/Investigational Product Accountability/Compliance; Collect Bottles/Atorvastatin Accountability/Compliance (for Week 10 and Week 14). |
| | | Added procedure "Hepatitis B Virus and Hepatitis C Virus Tests" at Screening Visit 1. |
| | | Transient Elastography timepoint added: ET/EOS. (Also, added this procedure to Section 9.7.15) |
| | | The list of assessments replaced with 3 broad subcategories: PD Assessments; Markers of Inflammation, Fibrosis, or Apoptosis; and Vitamin D. |
| | | Added footnote l to Serum Chemistry |
| | <del>Urine Based β-hCG-</del> Pregnancy Test <sup>q</sup> | Pregnancy Test <sup>q</sup> |
| | | Added hepatitis B and hepatitis C tests at Screening Visit 1 |
| | <sup>d</sup> Heart rate, blood pressure, temperature, and respiratory rate | <sup>d</sup> <b>Sitting</b> heart rate, blood pressure, temperature, and respiratory rate |

| Section | Original Text (Original protocol) | | | Revised Text (Ver | sion 2) | |
|---|---|---|---|---|---|---|
| | <sup>n</sup> Serum samples will be collected for lipoprotein analyses | | | <sup>n</sup> Serum <b>and plas</b><br>analyses | <sup>n</sup> Serum <b>and plasma</b> samples will be collected for lipoprotein analyses | |
| | [BNP]). s At selected investigational sites, subjects will have the option to provide blood samples for measurement of OCA PK. | | | β-hCG pregnancy | <sup>q</sup> Serum pregnancy test will be administered if urine-based β-hCG pregnancy test is positive. <b>Screening pregnancy tests will be serum-based tests.</b> | |
| | | | | plasminogen acti | <sup>r</sup> <b>Includes</b> markers of cardiovascular risk (adiponectin, plasminogen activator inhibitor-[(PAI-1], and B-type natriuretic peptide [BNP]). | |
| | | | | s At selected investigational sites, subjects will have the option to provide blood samples for measurement of OCA PK. PK samples will be collected within 30 minutes prior to dosing and again at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until the 1 hour sample is collected. | | |
| 7.1 | Header row updated as follows | | | | | |
| Overall Study Design (Table 2) | Month 3 | Month 6 | Month 9 | Month 3,<br>Month 15 | Month 6,<br>Month 18 | Month 9,<br>Month 21 |
| | | | | | Markers of Inflamm | 3 broad subcategories:<br>nation, Fibrosis, or |
| | | | | Additional timepoints added as follows: AUDIT alcohol measures: EOS/ET (Also, added this procedure to Section 9.7.20.) | | |
| | | | | Timepoints remo<br>Reverse Choleste<br>Month 15, and M | rol Transport analy. | sis: Month 3, Month 9, |

|---|---|---|
| | <sup>d</sup> Heart rate, blood pressure, temperature, and respiratory rate. | <sup>d</sup> <b>Sitting</b> heart rate, blood pressure, temperature, and respiratory rate. |
| | | <sup>1</sup> NOTE: Any time atorvastatin is up-titrated or reinitiated, a telephone safety contact must be conducted to assess AEs, concomitant medications, and atorvastatin compliance. |
| | | All subsequent footnotes have been adjusted by one |
| 7.4.2 | | Added: |
| Atorvastatin Dose<br>Adjustments | | If at any time during the double-blind or LTSE phases, serum chemistry results indicate LDLc <40 mg/dL, the subject should be brought back to the site within 1 to 2 weeks after the first result is obtained for an unscheduled (repeat) laboratory assessment. If LDLc <40 mg/dL is obtained on 2 consecutive visits, the subject may discontinue or reduce the dose of atorvastatin. |
| | | Subjects may also interrupt or discontinue atorvastatin due to tolerability issues including muscle-related symptoms (Section 5.8) and abnormal liver biochemistry. Any muscle-related complaints should be assessed per the ACC/AHA Guidelines (Appendix A) and statin dose adjusted accordingly: |
| | | • To avoid unnecessary discontinuation of statins, obtain a history of prior or current muscle symptoms to establish a baseline prior to initiation of statin therapy. |
| | | • If mild to moderate muscle symptoms develop during statin therapy: |


|---|
| <ul> <li>Discontinue the statin until symptoms can<br/>be evaluated.</li> </ul> |
| <ul> <li>Evaluate the patient for other conditions<br/>that might increase the risk for muscle<br/>symptoms.</li> </ul> |
| <ul> <li>If muscle symptoms resolve, and if no<br/>contraindication exists, re-challenge the<br/>subject with the same or a reduced dose of<br/>atorvastatin to establish a causal<br/>relationship between the muscle symptoms<br/>and statin therapy.</li> </ul> |
| <ul> <li>Once a low dose statin is tolerated, the<br/>dose may be gradually increased as<br/>tolerated and clinically indicated.</li> </ul> |
| <ul> <li>If after 2 months without statin treatment,<br/>muscle symptoms or elevated CPK levels<br/>do not completely resolve, consider other<br/>causes of muscle symptoms.</li> </ul> |
| <ul> <li>If persistent muscle symptoms are<br/>determined to arise from a condition<br/>unrelated to statin therapy, or if the<br/>predisposing condition has been treated,<br/>resume statin therapy at the original dose.</li> </ul> |
| If unexplained severe muscle symptoms or fatigue<br>develop during statin therapy, discontinue the<br>statin and address the possibility of<br>rhabdomyolysis by evaluating CPK and |

|---|---|---|
| | | creatinine, and performing urinalysis for myoglobinuria. |
| | | Elevations in liver biochemistry should be monitored per protocol subject withdrawal criteria (Section 8.4 and Appendix B). |
| | | Subjects who discontinue atorvastatin may continue on investigational product through the double-blind and LTSE phases, as deemed appropriate by the Investigator and Medical Monitor, and provided they continue to meet exclusion criteria #4 (LDL <200 mg/dL). |
| 8.1<br>Subject<br>Population | Approximately 80 subjects with biopsy-confirmed NASH without evidence of hepatic decompensation who meet eligibility criteria will be enrolled at approximately 30 investigational sites in the US with experience in treating patients with NASH. | Approximately 80 subjects with biopsy-confirmed NASH without evidence of hepatic decompensation who meet eligibility criteria will be enrolled at approximately 30 investigational sites in the US. |
| 8.4<br>Subject<br>Withdrawal | Subsections were rearranged as follows: 8.4.1 Reasons for Mandatory Discontinuation of Investigational Product | 8.4.1 Reasons for Mandatory Discontinuation of Investigational Product or Atorvastatin |
| Criteria | 8.4.1.1 Pregnancy 8.4.1.2 Severe Drug-Induced Liver Injury 8.4.1.3 Clinical Laboratory Values | 8.4.1.1 Adverse Events ≥Grade 3 in Severity and Possibly, Probably, or Definitely Related to Investigational Product |
| | 6.4.1.5 Chilical Euboratory Variets | <b>8.4.1.2</b> Pregnancy |
| | | <b>8.4.1.3</b> Severe Drug-Induced Liver Injury |
| | | 8.4.1.4 Myonecrosis |
| | | 8.4.2 Reasons for Mandatory Interruption of Investigational Product |
| | | 8.4.2.1 Adverse Events ≥Grade 4 in Severity and Not or Unlikely Related to Investigational Product |
| | | 8.4.2.2 Suspected Mild or Moderate Drug-Induced Liver Injury |

|---|---|---|
| | 8.4.2—Other Reasons for Study or Treatment Discontinuation of Subjects | <b>8.4.3</b> Other Reasons for Study or Treatment Discontinuation of Subjects |
| | 8.4.3 Subject Discontinuation Notification | <b>8.4.4</b> Subject Discontinuation Notification |
| 8.4.1.1 Adverse Events ≥Grade 3 in Severity | | If a subject experiences an AE that is ≥Grade 3 in severity (Section 12.1.4) that is considered possibly, probably, or definitely related to investigational product, the investigational product must be discontinued. |
| 8.4.1.2<br>Pregnancy | Whenever the site is notified of a possible pregnancy, the subject should be asked to come in for an unscheduled visit to perform a serum pregnancy test. If a female subject becomes pregnant, the subject must stop taking investigational product immediately and be withdrawn from the study. The subject must be followed by the Investigator through pregnancy outcome. The mother (and infant) will be followed as considered appropriate by the Investigator and the Medical Monitor. For reporting purposes, pregnancy is not considered an AE. | Whenever the site is notified of a possible pregnancy, the subject should be asked to come in for an unscheduled visit to perform a serum pregnancy test. If a female subject becomes pregnant, she must discontinue treatment with investigational product and atorvastatin immediately, but should continue with the study visit schedule and must be followed by the Investigator through pregnancy outcome. The mother (and infant) will be followed as considered appropriate by the Investigator and the Medical Monitor. As described in Section 12.1.8.1, pregnancy is not considered an AE for reporting purposes. |
| 8.4.1.3 Severe Drug-Induced Liver Injury (Paragraph 2) | Subjects should be encouraged to continue study visits despite stopping investigational product for continued study data collection but may withdraw consent at any time. | Subjects who discontinue due to significant drug-induced liver injury must be followed until the AE has resolved, stabilized, or is not of clinical concern. |
| 8.4.1.4 | | Moderate myonecrosis as defined by creatine kinase ≥10x |
| Myonecrosis | | the untreated baseline levels or ULN. Muscle-related symptoms that do not necessitate mandatory discontinuation of investigational product or atorvastatin are detailed in Section 5.8. |
| 8.4.2.1<br>Adverse Events | | If a subject experiences an AE categorized as ≥Grade 4 in severity and not or unlikely related to investigational |

|---|---|---|
| ≥Grade 4 in Severity and | | product, at least a mandatory interruption of investigational product is required. |
| 8.4.2.2<br>Suspected Mild<br>or Moderate<br>Drug-Induced<br>Liver Injury | Deleted Section 8.4.1.3. (Clinical Laboratory Values) of the Original Protocol, and replaced with Section 8.4.2.2 (new text shown in the right column). Development of the following clinical laboratory values during the course of the double-blind and LTSE phases of the study mandates investigational product discontinuation: *An aminotransferase (aspartate aminotransferase [AST] or ALT) elevation that is > 3x ULN/baseline/nadir, or *Total bilirubin >1.5 mg/dL (25.7 µmol/L) AND >2x the predose value (average of all pretreatment values), or *When myopathy is diagnosed or suspected (confirm with CPK prior to permanent discontinuation; discontinue if CPK >10x ULN) Note: The mean of all Screening and Baseline values constitute the predose values. If a subject is required to discontinue investigational product due to an increase in aminotransferase or bilirubin, the subject must be followed at appropriate intervals until these parameters have returned to within the normal range or prestudy values, and/or are stable, or there is no ongoing clinical concern. | Because transient fluctuations of ALT or AST are common, and progression to severe drug-induced liver injury or acute liver failure is uncommon, automatic discontinuation of investigational product with an elevation of ALT or AST that is >3x ULN/baseline/nadir or total bilirubin >2x ULN/baseline/nadir, as described in Appendix B, may be unnecessary. If a subject develops signs of a mild or moderate event of drug-induced liver injury, regardless of causality, investigational product should be interrupted until the event has resolved or returned to baseline, but the subject should continue with the study visit schedule. The subject may restart treatment after resolution of the event or return to baseline. Follow-up procedures, including laboratory evaluations and physical examinations, must be performed after a maximum of 2 weeks of re-treatment and may be conducted at a local clinic if the subject is unable to return to the site. Results must be reported immediately to the site so the Investigator can determine if the subject will be allowed to continue treatment. |
| 9.2.<br>Concomitant<br>Medications | Relevant information about all concomitant medications (including prescribed, over-the-counter, or herbal preparations) taken prior to (ie, within 30 days of Day 1) and during the study must be recorded in the source documents and eCRF, as well as any dose or dose regimen changes that occur during the study. | Relevant information about all concomitant medications (including prescribed, over-the-counter, or herbal preparations) taken prior to (ie, within 12 months of Day 1) and during the study must be recorded in the source documents and eCRF, as well as any dose or dose regimen changes that occur during the study. |
|---|---|---|
| 9.2.3<br>Management of<br>Changes in<br>Cholesterol | During the double-blind phase of the study, the dose of atorvastatin administration should be as described in this protocol through Week 12. At the Week 12 Visit, Investigators may increase or decrease the dose of atorvastatin as clinically indicated. | During the double-blind phase of the study, the dose of atorvastatin administration should be as described in this protocol through Week 12 unless tolerability issues develop as referenced in Section 7.4.2. At the Week 12 Visit, Investigators may increase or decrease the dose of atorvastatin as clinically indicated. |
| 9.2.4 Prohibited Medications <u>And</u> Table 3 | •Prohibited throughout the double-blind phase of the study: | Prohibited throughout the double-blind phase of the study: Medications contraindicated in the atorvastatin label, including HIV and Hepatitis C protease inhibitors, clarithromycin, and itraconazole (refer to atorvastatin prescribing information in Appendix E for complete list). These medications are also prohibited during the LTSE phase if the subject continues to receive atorvastatin during the LTSE. |
| | | Note: These medications were also added to Table 3. |
| 9.4.2<br>Emergency<br>Unblinding<br>Procedures | The <del>DSMC</del> (refer to Section 13.8) will have access to the IWRS and will be able to unblind individual subjects. The <del>DSMC</del> will be provided aggregate data to review during closed sessions. | The <b>DMC</b> (refer to Section 13.8) will have access to the IWRS and will be able to unblind individual subjects. The <b>DMC will review aggregate data</b> during closed sessions. |
| 9.6.1<br>Fasting<br>Requirements at<br>Study Visits | All subjects must have been fasting for at least 8 hours prior to Screening Visit 2 (Week -1 Visit) and all subsequent study visits, as all analytes will be assayed in fasting blood or plasma samples (Table 1 and Table 2). | All subjects must have been fasting for at least 8 hours prior to Screening Visit 2 (Week -1 Visit) and all subsequent study visits, as all analytes will be assayed in fasting blood, <b>serum</b> , or plasma samples (Table 1 and Table 2). |
| 9.6.2<br>Grapefruit and<br>Grapefruit Juice | Grapefruit and grapefruit juice consumption should be discouraged following initiation of atorvastatin (please refer to atorvastatin prescribing information [reference: Appendix A]). | Grapefruit and grapefruit juice consumption should be discouraged following initiation of atorvastatin due to possible increases in plasma concentration of atorvastatin (please refer to atorvastatin prescribing information [Appendix E]). |

|---|---|---|
| 9.7.1<br>Visit Windows | The Week -1 Visit should occur within ±1 days of the visit day. | The Week -1 Visit should occur within ±1 days of the Randomization/Day 1 Visit. |
| | | (A row added to in-text table) |
| | | Week 6, Week 10, and Week 14 ±4 days (Contact visits) |
| 9.7.3<br>Screening Visit 1<br>Procedures | Subjects who are statin free (ie, no statin use within 4 weeks of Screening) must return for fasted serum chemistry labs and may proceed to the Randomization/Day 1 Visit once screening labs are available and eligibility is confirmed; subjects who need to wash out statin therapy are required to have a Week -1 Visit 4 weeks after Screening Visit 1. •Record prior (if within 6 months of Day 1) and current concomitant medications. | Subjects who are statin free (ie, no statin use within 4 weeks of Screening) must return for fasted serum chemistry labs at |
| | | hepatitis C antibody (and positive HCV ribonucleic acid [RNA]) testing to confirm study eligibility. |
| | •Perform a urine-based β-hCG pregnancy test for female subjects of childbearing potential. Perform serum pregnancy test in females of childbearing potential, if urine β-hCG pregnancy test is positive. | •Perform serum pregnancy test in females of childbearing potential. |
| 9.7.5.<br>Randomization/D<br>ay 1 Visit<br>Procedures | •Record prior (within 30 days of Day 1) and current concomitant medications. | •Record prior (since Screening Visit 1) and current concomitant medications. |
| 9.7.5 | Serial blood samples will be obtained for measurement of OCA and its conjugates prior to dosing and at 0.5, 0.75, 1, | Serial blood samples will be obtained for measurement of OCA and its conjugates <b>30 minutes</b> prior to dosing and at |

|---|---|---|
| Additional Day 1 Procedures for PK Subjects <u>And</u> 9.7.13.1 Additional Week 16 Procedures for PK Subjects | 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until the 4-hour sample is collected. Lunch will be provided following collection of the 4-hour PK sample; the lunch will be a meal replacement drink with nutrition information that has been submitted to and approved by the Sponsor in advance. | 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until the <b>1-hour</b> sample is collected. <b>Meal</b> will be provided following collection of the <b>1-hour</b> PK sample; the lunch will be a meal replacement drink with nutrition information that has been submitted to and approved by the Sponsor in advance. |
| 9.7.5<br>Randomization/D<br>ay 1 Visit<br>Procedures<br><u>And</u><br>Sections 9.7.7,<br>9.7.9, 9.7.11,<br>9.7.13, 9.7.15,<br>9.7.18, 9.7.19,<br>9.7.20 | – Plasma bile acids, 7α hydroxy 4 cholesten 3 one (C4), and FGF-19; serum IL-6, cytokeratin-18 neoepitope M30 (CK-18-M30), high-sensitivity C-reactive protein (hs-CRP), TNF-α, and Vitamin D; and markers of glucose metabolism (C-peptide, insulin, fasting plasma glucose, and HbA1c) | <ul> <li>PD assessments; markers of inflammation, fibrosis and apoptosis; and markers of glucose metabolism (see Table 4 and Table 9)</li> <li>Vitamin D</li> </ul> |
| 9.7.8 (Week 6 Safety Contact) <u>And</u> 9.7.10 (Week 10 Safety Contact) <u>And</u> 9.7.12 (Week 14 Safety Contact) | Note: The numbering of 9.7 subsections is changed in Version 2 compared to that in the Original protocol from Section 9.7.9 onwards due to the addition of new Subsections 9.7.8, 9.7 10, and 9.7.12. | This is a telephone contact with the subject to Review and record AEs Review and record concomitant medications Assess investigational product and atorvastatin compliance |

|---|---|---|
| 9.7.18<br>LTSE Month 3,<br>Month 6, Month<br>9, Month 15,<br>Month 18, and<br>Month 21 Visit<br>Procedures | •Perform a physical examination (only at Month 3 Visit). | •Perform a physical examination (only at Month 3 and Month 15 Visits). |
| (Section 9.7.15 of<br>Original<br>Protocol) | •Determine alcohol consumption (using AUDIT questionnaire [only at Month 6 Visit]). | •Determine alcohol consumption (using AUDIT questionnaire [only at Month 6 and Month 18 Visits]). |
| | •Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability. | •Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability. |
| | | <ul> <li>NOTE: If atorvastatin dose is up-titrated or re- initiated after dose interruption, a telephone safety contact must be conducted 2 weeks following the change in dose to assess for AEs, concomitant medications, and investigational product and atorvastatin compliance.</li> </ul> |
| | •Obtain blood samples for: | •Obtain blood samples for: |
| | - Lipoprotein analyses <del>and</del> reverse cholesterol | <ul> <li>Lipoprotein analyses</li> </ul> |
| | transport analytes | <ul> <li>Reverse cholesterol transport analytes (only at<br/>Month 6 and Month 18 Visits)</li> </ul> |
| 9.7.20<br>LTSE End of<br>Study/Early<br>Termination<br>Procedures | | •Determine alcohol consumption (using AUDIT questionnaire). |
| 9.7.21<br>Unscheduled<br>Safety Visits | An increase in aminotransferases (ALT or AST) to >3× baseline (and >ULN) or total bilirubin >2× baseline (and >ULN) should be followed by repeat testing within 48 to 72 hours of the serum chemistry to confirm the | An increase in aminotransferases (ALT or AST) to >3× baseline (and >ULN) or total bilirubin >2× baseline (and >ULN) should be followed by repeat testing within 48 to 72 hours of the serum chemistry to confirm the abnormalities |

|---|---|---|---|
| | , | | and to determine if they are increasing or decreasing (Appendix B). |
| 10.5<br>Atorvastatin<br>Tablets | | | Atorvastatin tablets for oral administration contain 10 mg, 20 mg, <b>and</b> 40 mg atorvastatin. |
| 10.5.3<br>Atorvastatin<br>Dispensation | clinically indicated. | | At subsequent visits, atorvastatin will be dispensed as clinically indicated. For doses higher than 20 mg, subject may take multiple atorvastatin tablets for a total dose of 40 mg or 80 mg, as clinically indicated. |
| 11.1 | (Deleted the following | g row) | |
| Efficacy<br>Assessments<br>(Table 4) | Bile acid synthesis and concentrations | C4 (7α hydroxy 4 cholesten 3 one), conjugated and unconjugated bile acids (possible) | |
| 11.1.1<br>Efficacy<br>Laboratory<br>Assessments | The complete list of planned laboratory assessments supporting primary, secondary, and exploratory objectives of the study is shown in Table 4, and includes parameters related to LDL metabolism, lipoprotein metabolism, reverse cholesterol transport, liver biochemistry and markers of liver function, markers of inflammation, glycemic control, and NASH disease severity marker CK-18-M30. | | The complete list of planned laboratory assessments supporting primary, secondary, and exploratory objectives of the study is shown in Table 4, and includes parameters related to LDL metabolism, lipoprotein metabolism, reverse cholesterol transport, liver biochemistry and markers of liver function, markers of inflammation, glycemic control, <b>OCA PD markers</b> , and NASH disease severity markers CK-18-M30 and CK-18-M65. |
| 11.1.2.1<br>Central Reading<br>of Liver<br>Histology | Kleiner <del>2012</del> | | Kleiner 2005 |
| Pharmacokinetic<br>and<br>Pharmacodynamic<br>Assessments | | | Added the following new subsection: 11.2.1 Pharmacodynamic Assessments |

|---|---|---|
| | 11.2.1. OCA, Bile Acids, and FGF-19 | Original subsection 11.2.1 is now 11.2.2. and is re-named as below |
| | | 11.2.2. Pharmacokinetic Assessments |
| 11.2.1.<br>Pharmacodynami<br>c Assessments | | 11.2.1. Pharmacodynamic Assessments PD assessments will be collected according to the Schedule of Study Procedures (Table 1 and Table 2) from all subjects to measure C4, FGF-19, and possibly conjugated and unconjugated bile acids (dependent on the results of the C4 and FGF-19 assessments). |
| 11.2.2 | 11.2.1. OCA, Bile Acids, and FGF-19 | 11.2.2. Pharmacokinetic Assessments |
| Pharmacokinetic<br>Assessments<br>(Paragraph 1) | Subjects who participate in the PK and/or PD assessment will provide blood samples for the measurement of OCA and its conjugates, C4, FGF-19, and possibly bile acids, prior to administration of investigational product (predose) on Day 1 and at the Week 16 Visit. | Subjects who <b>opt to</b> participate in the PK assessment will provide blood samples for the measurement of OCA and its conjugates. <b>The first sample should be collected within 30 minutes</b> prior to administration of investigational product (predose) on Day 1 and at the Week 16 Visit. |
| Pharmacokinetic<br>Assessments<br>(Paragraph 2) | Instructions regarding the number and type of samples, including the PK assessments, to be collected at each visit, the required sample volumes, sample collection methods, sample processing, labeling, and shipping will be provided in a study specific laboratory manual. All necessary collection supplies will be provided by the central laboratory and will be appropriately assembled for the specific evaluations required at each visit. | |
| 12.1.8.1<br>Pregnancy and<br>Follow-Up | Pregnancies are not considered AEs in and of themselves; however, if a female study participant becomes pregnant while she is enrolled in the clinical study, she must discontinue treatment with investigational product immediately (see Section 8.4.1.1) and the Sponsor must be | Pregnancies are not considered AEs in and of themselves; however, if a female study participant becomes pregnant while she is enrolled in the clinical study, she must discontinue treatment with investigational product and atorvastatin immediately (see Section 8.4.1.1) and the |

|---|---|---|
| | notified within 24 hours of the Investigator's learning of the pregnancy by completing the Pregnancy Report eCF in the EDC system. | Sponsor must be notified within 24 hours of the Investigator's learning of the pregnancy by completing the Pregnancy Report eCRF in the EDC system. |
| | Women who discontinue the study due to pregnancy manot re-enroll in the study at any point. | Women who discontinue the study due to pregnancy may not re-enroll in the study at any point, but should continue with the study visit schedule and must be followed by the Investigator through pregnancy outcome. |
| 12.2.6<br>Laboratory<br>Assessments<br>(Table 9) | Serum chemistry Albumin, BUN, creatinine, conjugated (direct) bilirubin, total bilirubin, AST, ALT, ALP, GGT, creatinine, electrolytes (calcium, chloride, magnesium, phosphorus, potassium, sodium), total protein, bicarbonate, free fatty acids; and blood lipids (total cholesterol, LDL, HDL, and VLDL fractions and TGs) | Serum chemistry Albumin, BUN, creatinine, conjugated (direct) bilirubin, total bilirubin, AST, ALT, ALP, GGT, creatine phosphokinase, electrolytes (calcium, chloride, magnesium, phosphorus, potassium, sodium), total protein, bicarbonate, free fatty acids; and blood lipids (total cholesterol, LDL, HDL, and VLDL fractions and TGs) |
| | | Hepatiti s virus hepatitis B surface antigen, hepatitis C antibody, and screenin HCV ribonucleic acid [RNA] |
| 13.6.3.8<br>Cardiovascular<br>Risk Scores | New Section 13.6.3.8 Added | The cardiovascular risk score includes the FRS and Reynolds scores. Each score is derived from a subject's age, sex, smoking status, total cholesterol and HDL levels, systolic blood pressure, and other factors including family history, BMI, ethnicity, and medications. Cardiovascular scores will be calculated at the time of data analysis. These markers will be summarized by treatment group using descriptive statistics at Baseline and at each onstudy evaluation. The change and percentage change from Baseline will also be summarized. |

|---|---|
| 13.9.<br>Adjudication<br>Committees | All suspected major adverse cardiovascular events (MACE), and drug-related hepatic injury events that occur after administration of the first dose of investigational product will be reviewed by the following blinded adjudication committees, depending on event type, before inclusion in any analysis. The 2 committees and event types they are responsible for adjudicating are as follows: |
| | •Cardiovascular Events Committee (CEC): Adjudicates all suspected MACE (Appendix D) |
| | •Hepatic Safety Committee: Adjudicates all suspected drug-related hepatic injury events |
| | Each adjudication committee will have a charter that documents the reporting of events by the study site; definition of the suspected events to be adjudicated; supply of source documentation to the committee; and the entire data flow and process from committee membership, review of the events by the committee, reporting of the final assessment, and the working procedures of the committee. |
| | The adjudication committee members will include experts with relevant adjudication experience; they will not be involved in the study as Investigators, DMC members, or consultants. Any candidate found to have a conflict or whose name is listed on the FDA debarment list will not be offered membership. Conflicts of interest are assessed regularly, and if members are found to have a new conflict of interest they will be replaced. |
| | The adjudication of suspected events will be based on available source documentation, including but not limited to individual clinical study data, hospital records, histology, discharge summaries, and/or death certificates. The adjudication committees will not receive any |

|---|---|
| | individual subject treatment or site-specific information. The assessment of events will be conducted in compliance with study-specific procedures, manuals, GCP, and all other applicable regulatory requirements, including the archiving of essential documents. |
| 19.<br>List of<br>References | American Diabetes Association. Standards of medical care in diabetes-2013. Diabetes Care. 2013;36(Suppl 1):S11-S66. |
| | Desai CS, Martin SS, Blumenthal RS. Non-cardiovascular effects associated with statins. BMJ 2014;349:g3743 |
| | Kleiner D, Brunt E, Van Natta M, et al. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology 2005;41:1313-1321. |
| | Mampuya WM, Frid D, Rocco M, et al. Treatment strategies in patients with statin intolerance: the Cleveland Clinic experience. Am Heart J. 2013;166:597-603. |
| | Rosenson RS, Baker SK, Jacobson TA et al. An assessment by the statin muscle safety task force: 2014 update. J Clin Lipid. 2014;8:S58-S71. |
| | Simic I, Reiner Z. Adverse effects of statins – myths and reality. Curr Pharm Des. 2015;21:1220-1226. |
| | Zhang H, Plutzky J, Skentzos S, et al. Discontinuation of statins in routine care settings: a cohort study. Ann Intern Med. 2013;158:526-534. |

Version 4: 19 Dec 2016 Protocol 747-209

|---|---|---|
| Appendix A | APPENDIX A. <del>EUROPEAN AND NICE</del> GUIDANCE<br>FOR THE USE OF STATINS | APPENDIX A. AMERICAN COLLEGE OF CARDIOLOGY/AMERICAN HEART ASSOCIATION GUIDANCE FOR THE USE OF STATINS |
| Appendix B | For subjects who progress to cirrhosis and decompensation while participating in the study, elevation in liver biochemistry and development of other laboratory and clinical abnormalities may be expected. Clinical outcomes should be reported and recorded as described in Section 12.1.5 and appropriate action should be taken regarding investigational product use and study participation as described in Section 8.4. | For subjects who progress to cirrhosis and decompensation while participating in the study, elevation in liver biochemistry and development of other laboratory and clinical abnormalities may be expected. Clinical adverse events (AEs) should be reported and recorded as described in Section 12.1.5 and appropriate action should be taken regarding investigational product use and study participation as described in Section 8.4. |
| | In subjects with abnormal ALT/AST or bilirubin at baseline, fold increase should be assessed against baseline levels instead of ULN as follows: 3× baseline ALT/AST (and >200 IU/L), or total bilirubin >2× baseline (and >2 mg/dL). | In subjects with abnormal ALT/AST or bilirubin at baseline, fold increase should be assessed against baseline levels instead of ULN as follows: 3× baseline ALT/AST, or total bilirubin >2× baseline (and >2 mg/dL). |
| Appendix D | | APPENDIX D. STANDARDIZED DEFINITIONS FOR CARDIOVASCULAR ENDPOINT EVENTS |

## APPENDIX G. 747-209 PROTOCOL VERSION 3 SUMMARY OF CHANGES

Protocol 747-209 was revised to add a modified randomization scheme to the LTSE in order to maintain the blind of the double-blind phase. The list of conjugates or metabolites of OCA for assessment was expanded to include OCA glucuronide. Additionally, various aspects of the study design and study population were clarified.

## **Summary of Changes**

The following revisions were made to the protocol in Protocol Version 3. Revised and new text in Version 3 is indicated in bold font, and the text deleted from Protocol Version 3 is crossed out in the table below. Minor/editorial changes are not listed individually in the summary table below.

| Section | | Original Text | | Revised Text |
|---|---|---|---|---|
| Global change | Oral temperature | | Body temperature | |
| Global change | OCA, tauro-OCA, glyco-OCA, total OCA, potentially other conjugates or metabolites not yet identified | | | glyco-OCA, total OCA, <b>OCA glucuronide</b> , njugates or metabolites not yet identified |
| Title Page | | Version 2: 22 October 2015 | | The CONTROL Study CA aNd STatin for MonitoRing Of Lipids Version 3: 14 June 2016 |
| Study Personnel<br>Contact<br>Information | Primary<br>Medical<br>Monitor<br>Contact:<br>Email: | Roya Hooshmand-Rad, MD, PhD<br>Executive Director, Clinical Research<br>Intercept Pharmaceuticals, Inc. (Intercept)<br>rhooshmand-rad@interceptpharma.com | | vidual medical monitors may also be the NASH medical monitor hotline and Emad Basta, MD (Lead) Medical Monitor/Medical Expert PRA Health Sciences +1 630 235 6201 CONTROL@PRAHS.com +1 844 250 6396 NASH209@interceptpharma.com |

| Section | Original Text | Revised Text |
|---|---|---|
| | | Email Secondary Roya Hooshmand-Rad, MD, PhD |
| | Secondary Barbara Scholz, MD Contact: Medical Director, Drug Safety | Contact: Executive Director, Medical Safety and Pharmacovigilance Intercept Pharmaceuticals, Inc. (Intercept) |
| | Intercept +1 858 353 1350 (Pacific time zone) | Mobile +1 858 880 6485 (Pacific time zone) Phone: rhooshmand-rad@interceptpharma.com Email: |
| | Email: barbara.scholz@interceptpharma.com | Barbara Scholz, MD Secondary Contact: Barbara Scholz, MD Medical Director, Drug Safety Intercept |
| | | Mobile Phone: Email: +1 858 353 1350 (Pacific time zone) barbara.scholz@interceptpharma.com |
| Synopsis Objectives, 6.3 Exploratory Objectives | To evaluate improvement in noninvasive-radiological assess of fibrosis via transient elastography (TE; at sites where availand evaluated at the end of LTSE) | |
| Synopsis<br>Methodology,<br>7.1 Overall Study | Statin-treated subjects will be required to stop statin treatment (after signing informed consent) for a total of 5 weeks prior transformation. | o (after signing informed consent) for <b>up to</b> 5 weeks, <b>including a 4-week statin washout period</b> , prior to <b>Randomization/Day1</b> . |
| Design | Screening Period: Subjects using statins within 30 days of the initial Screening (Screening Visit 1) are required to stop statin therapy immed following this initial visit and must undergo a 4-week statin washout period. One week prior to randomization (Screenin Visit 2; Week 1), these subjects will have a pre-randomizati visit for assessment of their fasting LDL cholesterol levels. | visit (Screening Visit 1) are required to stop statin therapy immediately following this initial visit and must undergo a 4-week statin washout period <b>prior to Screening Visit 2</b> . At |

| Section | Original Text | Revised Text |
|---|---|---|
| | Subjects with fasting LDL cholesterol values >200 mg/dL at Week 1 will be excluded from the study and their NASH should be managed according to standard of care. | Subjects with fasting LDL cholesterol values >200 mg/dL at Screening Visit 2 will be excluded from the study and their dyslipidemia should be managed according to standard of care. |
| | Double Blind: | Double Blind: |
| | Subjects who discontinue atorvastatin during the double-blind phase are eligible to continue OCA during the double-blind phase and enroll into the LTSE at the discretion of the Investigator, provided they continue to meet exclusion criteria #4 (LDL <200 mg/dL). | Subjects who discontinue atorvastatin during the double-blind phase are eligible to continue OCA during the double-blind phase and enroll into the LTSE at the discretion of the Investigator, provided they continue to meet <b>the LDLc cutoff of</b> exclusion criteria #4 ( <b>ie</b> , LDL <b>c</b> <200 mg/dL). |
| | LTSE Phase: | LTSE Phase: |
| | During the LTSE phase, all subjects will be treated with OCA. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will receive OCA 10 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg with no tolerability concerns will titrate to OCA 25 mg. Subjects who are randomized to the OCA 25 mg treatment group will continue receiving OCA 25 mg during the LTSE. | During the LTSE phase, all subjects will be treated with open-label OCA 10 mg or OCA 25 mg. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will be randomized in a 1:1 ratio to receive OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg or OCA 25 mg during the double-blind phase will continue on the same dose throughout the LTSE. |
| Synopsis<br>Methodology,<br>7.1.1 Study<br>Design | Placebo Statin Vashout Placebo Statin Vashout Placebo 10 mg OCA Statin Vashout Placebo 10 mg OCA 25 mg OCA Quarterly Visits* *Subjects initiating the LTSE are required to have a safety contact 4 weeks into the LTSE | Randomization Double-Blind Treatment Period Statin Statin Titrated Statin use per EU/US Guidelines Placebo Screening & Statin Use per EU/US Guidelines Placebo 10 mg OCA Statin Use per EU/US Guidelines Placebo 10 mg OCA 25 mg OCA Quarterly Visits Wk -5 Wk Wk 4 Wk 8 Wk 12 Wk 16 LTSE Wk 4 |
| Synopsis Number of Subjects, 7.2 Number of Subjects | 8. At least 67% (n = 54) of subjects enrolled in the study will have fibrosis stage 1 and up to 33% (n = | 9. A maximum of 20% of subjects will have stage 4 fibrosis. |

**Original Text Revised Text** Section 26) of subjects will have fibrosis stage 2, stage 3, or stage 4 Synopsis, Key 6. Contraception: Female subjects of childbearing 6. Contraception: Female subjects of Inclusion Criteria potential must use ≥1 effective method of childbearing potential must use ≥1 effective 8.2 Subject contraception during the study and until 30 days method of contraception during the study and Inclusion Criteria following the last dose of investigational until 30 days following the last dose of product. Effective methods of contraception investigational product. Effective methods of are considered to be those listed below. contraception are considered to be those listed below <del>Double-barrier method, ie, (a) condom (male or</del> female) or (b) diaphragm, with spermicide Barrier method, ie, condom (male or female) with spermicide or diaphragm with spermicide Intrauterine device Intrauterine device Vasectomy (partner) Vasectomy (partner) Hormonal (eg., contraceptive pill, patch, intramuscular implant or injection) Hormonal (eg, contraceptive pill, patch, intramuscular implant or injection) Abstinence (defined as refraining from heterosexual intercourse) Abstinence (defined as refraining from heterosexual intercourse) Synopsis, Key 8 Uncontrolled diabetes defined as HbA1c>9 0% 8. Uncontrolled diabetes defined as Exclusion within 60 days prior to randomization (Day 1). HbA1c≥9.5% within 60 days prior to Criteria 9. Administration of any of the following randomization (Day 1) 8.3 Subject medications as specified below: Exclusion 9. Administration of any of the following Criteria Prohibited 30 days prior to Day 1: medications as specified below: - bile acid sequestrants including cholestyramine Prohibited 30 days prior to Day 1: Prohibited 3 months prior to Day 1: bile acid sequestrants including nicotinic acid and derivatives, ezetimibe, or cholestyramine, and its derivatives any prescription or over-the-counter medication or herbal remedy with putative NASH efficacy Prohibited 3 months prior to Day 1: (except Vitamin E or TZDs), nicotinic acid and derivatives, ezetimibe, or fenofibrate or other fibrates, or

| Section | Original Text | Revised Text |
|---|---|---|
| | <ul> <li>Any over-the-counter or health foods used to<br/>treat lipids including plant sterols and berberine</li> </ul> | <ul> <li>any prescription or over-the-counter<br/>medication or herbal remedy with putative<br/>NASH efficacy (except Vitamin E or TZDs),<br/>or</li> </ul> |
| | <ul> <li>10. Evidence of other forms of chronic liver disease including but not limited to:</li> <li>Positive test result at Screening for hepatitis B surface antigen or hepatitis C antibody (and positive hepatitis C virus [HCV] ribonucleic acid [RNA])</li> <li>Primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis or overlap syndrome</li> <li>Alcoholic liver disease</li> <li>Wilson's disease or hemochromatosis or iron overload as defined by presence of 3+ or 4+ stainable iron on liver biopsy</li> <li>Alpha-1-antitrypsin (A1AT) deficiency as defined by diagnostic features in liver histology (confirmed by A1AT level less than normal; exclusion at the Investigator's discretion)</li> </ul> | <ul> <li>ursodeoxycholic acid, or</li> <li>fenofibrate or other fibrates, or</li> <li>Any over-the-counter or health foods used to treat lipids including plant sterols and berberine</li> <li>Evidence of other forms of known chronic liver disease including but not limited to: <ul> <li>Positive test result at Screening for hepatitis B surface antigen</li> </ul> </li> <li>Active hepatitis C virus (HCV) infection (positive for HCV ribonucleic acid [RNA] at Screening) or history of positive HCV RNA test result</li> <li>Primary biliary cirrhosis (also known as primary biliary cholangitis), primary sclerosing cholangitis, autoimmune hepatitis or overlap syndrome</li> </ul> |
| | <ul> <li>Prior known drug-induced liver injury within 5 years before Day 1</li> <li>Known or suspected hepatocellular carcinoma</li> <li>17. Platelet count &lt;100,000/mm³ at any Screening Visit</li> <li>24. Receipt of any investigational product not being</li> </ul> | <ul> <li>Alcoholic liver disease</li> <li>Wilson's disease or hemochromatosis or iron overload as defined by presence of 3+ or 4+ stainable iron on liver biopsy</li> <li>Alpha-1-antitrypsin (A1AT) deficiency as defined by diagnostic features in liver histology (confirmed by A1AT level less than normal; exclusion at the</li> </ul> |
| | evaluated for the treatment of diabetes or NASH within 30 days prior to Day 1 or within 5 half-lives of the compound (whichever was longer) before Day 1 | Investigator's discretion) |

| Section | | | Original Text | | | | Revised Text |
|---|---|---|---|---|---|---|---|
| | | | | | | | own drug-induced liver injury within before Day 1 |
| | | | | | • Kr | nown o | or suspected hepatocellular carcinoma |
| | | | | | 17. Pla | atelet c | count <75 000/mm³ at any Screening Visit |
| | | | | | ev<br>fre<br>pri<br>co | aluated<br>om Sci<br>ior to I<br>mpoun | of any investigational product not being d for the treatment of diabetes or NASH reening Visit 1 to Day 1, within 30 days Day 1, or within 5 half-lives of the nd before Day 1 (whichever was longer) holecystitis or acute biliary obstruction |
| Synopsis,<br>Duration of<br>Subject<br>Participation | | | statin-using subjects: 4-week statin reening (5-weeks (statin-using subjects | | | | r statin-using subjects: Up to 5 weeks k statin washout period) |
| Synopsis, Criteria | Exploratory Endpoints | | | Exploratory I | Endpoi | ints | |
| for Evaluation 11.1 Efficacy Assessments, Table 4 | OCA<br>pharmacokinet | tics | OCA, tauro-OCA, glyco-OCA, total OCA, potentially other conjugates or metabolites not yet identified | | OCA<br>pharmacokinet | tics | OCA, tauro-OCA, glyco-OCA, total OCA, <b>OCA glucuronide</b> , potentially other conjugates or metabolites not yet identified |
| | Noninvasive<br>radiological liv<br>fibrosis<br>measurements | ver | By TE (where available <del>, and evaluated at the end of LTSE</del> ) | | Noninvasive radiological liv fibrosis measurements | | By TE (where available) |
| List of | PBC | nrimo | ry biliary cirrhosis | | PBC | | ary biliary <b>cholangitis (also known as</b> |
| Abbreviations | 1 BC | prima | 1 y Ulliat y Cliffiusis | $-\parallel$ | 1 BC | | nary biliary cirrhosis) |
| and Definitions<br>of Terms | | | | | CAC | | diovascular Adjudication<br>nmittee |

| Section | Original Text | Revised Text |
|---|---|---|
| 5.5 Clinical<br>Experience with<br>Obeticholic Acid | OCA is under investigation for the treatment of multiple chronic liver diseases, including the treatment of NASH, primary biliary cirrhosis (PBC), primary sclerosing cholangitis (PSC), and biliary atresia. The clinical development program for OCA includes the following 3 studies conducted using subjects with NAFLD or NASH: " | OCA is under investigation for the treatment of multiple chronic liver diseases, including the treatment of NASH, primary biliary cholangitis (PBC, also called primary biliary cholangitis (PBC, also known as primary biliary cirrhosis [Beuers 2015a, Beuers 2015b, Beuers 2015c]), primary sclerosing cholangitis (PSC), and biliary atresia. The clinical development program for OCA includes the following 3 studies conducted using subjects with NAFLD or NASH: |
| | Study D8602001: An ongoing Phase 2 study being conducted by Intercept's development partner (Sumitomo Dainippon Pharma Co., Ltd) to evaluate the efficacy and safety of 3 doses of OCA versus placebo in NASH. | Study D8602001: A Phase 2 study conducted by<br>Intercept's Asian development partner (Sumitomo<br>Dainippon Pharma Co., Ltd) to evaluate the efficacy and<br>safety of 3 doses of OCA versus placebo in NASH |
| | Study D8602001 is ongoing and remains blinded. | Study D8602001 demonstrated a dose-dependent increase in the percentage of OCA-treated subjects compared to placebo subjects who achieved the primary endpoint (p = 0.053, not significant). The 40 mg OCA dose group achieved statistical significance for the primary endpoint compared to placebo (p = 0.0496). Dose-dependent trends not reaching statistical significance were also observed for several other prespecified histologic endpoints, including the proportion of subjects with steatosis and inflammation improvement, ballooning resolution, and NASH resolution. In the completer analysis, similar dose-dependent effects were observed, with 51% of patients in the 40 mg dose group compared to 22% in the placebo group meeting the primary endpoint (p = 0.0061). With the exception of dose-dependent pruritus, OCA appeared to be generally safe and well tolerated. The number of pruritus-associated discontinuations were 0, 0, 2, and 5 subjects in the placebo, 10 mg, 20 mg, and 40 mg OCA groups, respectively. Changes in lipid parameters were directionally similar to those observed in the FLINT study. No other meaningful differences in the rate of AEs between the OCA and placebo groups were noted. |

| Section | Original Text | Revised Text |
|---|---|---|
| 5.6.6 Rationale<br>for Timing of<br>Unblinding<br>Process and<br>Implications in<br>LTSE | For those subjects continuing into the LTSE: Following completion of all study procedures associated with the double-blind period, subjects will be unblinded via the interactive web response system (IWRS) to determine the open label OCA dose to be initiated in the LTSE. This will allow double blind, placebo-treated subjects to initiate OCA at an appropriate dose, and OCA-treated subjects to maintain or increase their dose based on therapeutic response and tolerability rather than forcing fixed dosing to maintain the blind. | As Study 747-209 is a randomized, double-blind study, the double-blind data will not be unblinded until all double-blind data are final and the database is locked. Accordingly, all subjects continuing in the LTSE, investigators, and the Sponsor will remain blinded to subjects' DB treatment regimen. Subjects who were receiving placebo or 5 mg OCA in the DB phase will be randomized to receive either OCA 10 mg or OCA 25 mg in the LTSE. Subjects who were receiving OCA 10 mg or OCA 25 mg in the DB phase will continue on the same dose throughout the LTSE. Using this approach, blinding of the trial will be maintained. |
| 5.8 Summary of<br>Known Potential<br>Risks with<br>Atorvastatin | | If treatment with statins is initiated, women of childbearing potential must be informed that statin use is contraindicated during pregnancy. Methods of contraception should be reviewed and modified, if necessary, to ensure highly effective methods with failure rates <1% per year, such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or history of vasectomy of partner are used. |
| 7.1.2 Schedule of<br>Study<br>Procedures,<br>Double-Blind<br>Period | <ul> <li><sup>a</sup> Subjects using statins within 4 weeks of Screening are required to stop administering statin therapy after Screening Visit 1, and must undergo a 5 week washout period prior to randomization.</li> <li><sup>b</sup> Screening Visit 2 is required for all subjects. All subjects must have been fasting for at least 8 hours prior to the visit. For subjects undergoing a 4-week washout period, this visit will occur at Week 1. For subjects not taking statins at Screening Visit 1, this visit can occur at any time after Screening Visit 1 and up to 1 week prior to randomization. For subjects</li> </ul> | Added Weeks row to clarify timing of Screening Visits Modified Visit windows for Screening Visit 1: Day -35 to Day -7 Modified Visit window for Screening Visit 2: Day -7 to Day -1 a Subjects using statins within 4 weeks of Screening are required to stop administering statin therapy after Screening Visit 1, and must complete a 4-week statin washout prior to performing assessments at Screening Visit 2. b Screening Visit 2 is required for all subjects. All subjects must have been fasting for at least 8 hours prior to the visit. The Randomization/Day 1 Visit may occur as soon as screening labs are available and eligibility is confirmed for all subjects. For subjects undergoing a 4-week washout period, Screening Visit 2 may occur on day 28 (±1) day of the washout period. For subjects not taking statins at Screening Visit 1, Screening Visit 2 can occur at any time |

| Section | Original Text | Revised Text |
|---|---|---|
| | using statins within 4 weeks prior to Screening Visit 1, Screening Visit 2 can occur at any time after 4 weeks have lapsed since the subject's last statin dose. | within 28 days after Screening Visit 1. All Screening assessments must be completed ≤35 days prior to the Randomization/Day 1 Visit. |
| | d Sitting heart rate, blood pressure, temperature, and respiratory rate i and none of the exclusion criteria, may be randomized." | <sup>d</sup> Sitting heart rate, blood pressure, <b>body</b> temperature, and respiratory rate |
| | <sup>k</sup> Blood samples for all analyses will be collected predose (before administering investigational product) on indicated visit days. | i and none of the exclusion criteria, may be randomized. Subjects randomized to placebo or OCA 5 mg during the double-blind period will be randomized to OCA 10 or 25 mg during the LTSE k Blood samples for all analyses will be collected predose (before administering investigational product or atorvastatin) on indicated visit days. |
| 7.1.2 Schedule of<br>Study<br>Procedures,<br>LTSE | a The first visit after start of LTSE (Month 1 Visit) is relative to Week 16 Visit of the double-blind phase (LTSE Day 1 Visit). This is not a study site visit. The subject should be contacted approximately 1 month after the start of the LTSE, and compliance with OCA treatment instructions, concomitant medications, and AEs should be assessed. d Sitting heart rate, blood pressure, temperature, and respiratory rate | <ul> <li>Month 1</li> <li>Added: <ul> <li>Fast ≥8 h Prior to Visit</li> <li>Vital Signs</li> <li>Collect Bottles/Atorvastatin</li></ul></li></ul> |
| 7.3 Treatment<br>Assignment | Eligible subjects will be randomized into 4 groups in a 1:1:1:1 ratio to receive OCA 5 mg, OCA 10 mg, OCA 25 mg, or placebo during the double-blind phase of the study. Randomization will | Eligible subjects will be randomized into 4 groups in a 1:1:1:1 ratio to receive OCA 5 mg, OCA 10 mg, OCA 25 mg, or placebo during the double-blind phase of the study. |

| Section | Original Text | Revised Text |
|---|---|---|
| | be stratified by LDL concentration (fasting serum LDL cholesterol at Screening Visit 2; $\leq$ 125 mg/dL or $>$ 125 mg/dL) and baseline fibrosis stage (stage 1, 2 or stage 3, 4). All subjects will also receive atorvastatin starting at Week 4 at 10 mg daily, escalating to 20 mg at Week 8 (if 10 mg daily is tolerated), with further dose adjustments to be performed as clinically indicated at Week 12, and throughout the LTSE phase. Subjects randomized to placebo or OCA 5 mg will receive OCA 10 mg during the LTSE; subjects randomized to OCA 10 mg or OCA 25 mg will receive OCA 25 mg during the LTSE. The study design schematic is shown in Figure 1. | Randomization will be stratified by LDL concentration (fasting serum LDL cholesterol at Screening Visit 2; ≤125 mg/dL or >125 mg/dL) and baseline fibrosis stage (stage 1, 2 or stage 3, 4). All subjects will also receive atorvastatin starting at Week 4 at 10 mg daily, escalating to 20 mg at Week 8 (if 10 mg daily is tolerated), with further dose adjustments to be performed as clinically indicated at Week 12, and throughout the LTSE phase. Subjects will receive open-label OCA 10 mg or OCA 25 mg during the LTSE depending on their double-blind randomized dose (see Section 7.1). The study design schematic is shown in Figre 1. |
| 7.4.1<br>Investigational<br>Product Dose<br>Adjustments | During the LTSE phase, all subjects will be treated with OCA. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will receive OCA 10 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg with no tolerability concerns will titrate to OCA 25 mg. Subjects randomized to OCA 25 mg will continue to receive this dose throughout the LTSE. Subjects may continue with atorvastatin therapy as clinically indicated. | During the LTSE phase, all subjects will be treated with OCA. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will be re-randomized in a 1:1 ratio through IWRS to OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg will continue to receive OCA 10 mg throughout the LTSE. Subjects randomized to OCA 25 mg will continue to receive OCA 25 mg throughout the LTSE. Subjects may continue with atorvastatin therapy as clinically indicated. |
| 8.4.1.3 Severe<br>Drug-Induced<br>Liver Injury | Subjects who develop significant drug-induced liver injury, which is considered to be causally related to the investigational product, should be discontinued from investigational product and should not be rechallenged. Significant injury as described in Appendix B, or evidence of functional hepatic impairment as indicated by rising bilirubin or INR. Natural progression of the underlying condition and other causal factors such as a common bile duct stone or development of other concurrent liver disease should be considered before the investigational product is permanently discontinued. Severe drug induced-liver injury that is not considered related to investigational product must be discussed with the Sponsor before resuming treatment. Subjects who discontinue due to significant drug-induced liver injury must be followed until the AE has resolved, stabilized, or is not of clinical concern. | If a subject develops signs and symptoms of a severe druginduced liver injury, regardless of causality, investigational product and atorvastatin should be interrupted until the event has resolved or returned to baseline, but the subject should continue with the study visit schedule. Subjects who develop significant drug-induced liver injury, which is considered to be causally related to the investigational product or atorvastatin, should be discontinued from investigational product or atorvastatin, as appropriate and should not be rechallenged. Significant injury as described in Appendix B, and includes evidence of functional hepatic impairment as indicated by rising bilirubin or INR. Natural progression of the underlying condition and other causal factors such as a common bile duct stone or development of other concurrent liver disease should be considered before the investigational product is permanently discontinued. |

| Section | Original Text | Revised Text |
|---|---|---|
| | | Severe drug induced-liver injury that is not considered related to investigational product or atorvastatin must be discussed with the Sponsor before investigational product or atorvastatin is reinitiated. Follow-up procedures for subjects resuming treatment, including laboratory evaluations and physical examinations, must be performed after a maximum of 2 weeks of re-treatment and may be conducted at a local clinic if the subject is unable to return to the site. Results must be reported immediately to the site so the Investigator can determine if the subject is to be allowed to continue treatment. Subjects who discontinue due to significant druginduced liver injury must be followed until the AE has resolved, stabilized, or is not of clinical concern. |
| 9.1 Investigational Product and Atorvastatin Treatment Regimen | The investigational products are either OCA or placebo. | While placebo, OCA, and atorvastatin are all study medications provided by the Sponsor, for the purposes of this protocol, investigational product refers to OCA or placebo, and study medication, where used, refers to atorvastatin. |
| 9.1.2 LTSE | Following completion of Week 16 Visit procedures, subjects who are participating in the LTSE will be unblinded via the IWRS. Subjects who were receiving OCA during the double blind phase will continue to receive either OCA 10 mg or OCA 25 mg once daily during the LTSE. Subjects randomized to placebo or 5 mg OCA during the double blind phase will initiate dosing at OCA 10 mg in the LTSE. Subjects randomized to OCA 10 mg during the double-blind phase will titrate to OCA 25 mg on Day 1 of the LTSE. Subjects randomized to OCA 25 mg during the double-blind phase will continue to receive OCA 25 mg. | Following completion of Week 16 Visit procedures, all subjects will be treated with open-label OCA 10 mg or OCA 25 mg. Subjects randomized to placebo or OCA 5 mg during the double-blind phase will be randomized in a 1:1 ratio to receive OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase. Subjects randomized to OCA 10 mg or OCA 25 mg during the double-blind phase will continue on the same dose throughout the LTSE. |
| 9.2.5 Standard of<br>Care and Other<br>Concomitant<br>Medications | Subjects taking BAS or aluminum hydroxide- or smectite-containing antacids should be instructed to stagger their dosing of investigational product, ensuring at least 4 hours between doses of the BAS and/or antacids and the investigational product (ie, BAS should be administered 4 hours before or 4 hours after investigational product administration). | Subjects taking BAS (including cholestyramine and its derivatives, colestipol, colesevelam, or other sequestrants) or aluminum hydroxide- or smectite-containing antacids should be instructed to stagger their dosing of investigational product, ensuring at least 4 hours between doses of the BAS and/or antacids and the investigational product (ie, BAS should be |

| Section | Original Text | Revised Text |
|---|---|---|
| | | administered 4 hours before or 4 hours after investigational product administration). |
| | | Taken concomitantly, OCA and warfarin may decrease INR, thus INR should be monitored and the dosage of warfarin adjusted, as needed, to maintain the target INR range. |
| | | The effect of OCA on drug metabolizing enzymes has been evaluated in both in vitro and clinical studies. The PK profile of caffeine, a sensitive CYP1A2 substrate, showed weak effect of OCA on CYP1A2. Based on these results, OCA may increase the exposure of narrow therapeutic index drugs that are substrates for CYP1A2, such as theophylline and tizanidine. |
| 9.4<br>Randomization<br>and Blinding | The Investigator or designee will be required to register the subject in the IWRS and may be prompted to provide patient data necessary to properly randomize and allocate the subject to treatment. A randomization number will be assigned and investigational product (OCA or placebo) dispensing information will be provided (eg, bottle numbers allocated) while maintaining the study blind. The subjects, Investigator, and study site staff will be blinded to the subject's treatment allocation during the subject's participation-in the double-blind phase of the study. | The Investigator or designee will be required to register the subject in the IWRS and may be prompted to provide patient data necessary to properly randomize and allocate the subject to treatment. A randomization number will be assigned and investigational product (OCA or placebo) dispensing information will be provided (eg, bottle numbers allocated) while maintaining the study blind. The subjects, Investigator, and study site staff will be blinded to the subject's treatment allocation in the double-blind phase of the study until all subjects have completed the double-blind phase of the study and the database locked. |
| | | In the LTSE phase, all subjects will be treated with open-label OCA 10 mg or OCA 25 mg: subjects randomized to placebo or OCA 5 mg during the double-blind phase will be randomized in a 1:1 ratio to receive OCA 10 mg or OCA 25 mg upon entry into and throughout the LTSE phase and subjects randomized to OCA 10 mg or OCA 25 mg during the double-blind phase will continue on the same dose throughout the LTSE. |
| 9.4.2 Emergency<br>Unblinding<br>Procedures | Randomization codes and corresponding treatment assignments will be made available to the Investigator for emergency use only through the IWRS system. When possible, the Medical Monitor | Randomization codes and corresponding treatment assignments will be made available to the Investigator and the Medical Monitor for emergency use only through the IWRS system. |

| Section | | Original Text | | Revised Text |
|---|---|---|---|---|
| | necessitates unblinding (in blinded treatment is necess the subject). If it is not residually in advance of unblinding, document the case in the state investigator should compremature unblinding of the unblinding or unblinding for unblinding a subject's the Investigator. Similarly blind for the purpose of every regulatory reporting purpose. | e event that a medical emergency e, in situations where knowledge of the sary for further medical management of asonable to inform the Medical Monitor the Investigator must promptly subject's source record. Subsequently, intact the Medical Monitor to explain any reatment assignment (eg, accidental due to a serious AE [SAE]). Procedures treatment will be provided separately to y, if the Medical Monitor breaks the valuating an emergent safety issue or for coses, the Medical Monitor will document ince the rationale, circumstances, and the about the unblinding. | event that a medical eme situations where knowled for further medical mana reasonable to inform the unblinding, the Investigathe subject's source reco should contact the Medic unblinding of treatment a unblinding due to a serio unblinding a subject's treatment to the Investigator. The Medical Contact the Investigator. | cal Monitor should be consulted in the rgency necessitates unblinding (ie, in dge of the blinded treatment is necessary gement of the subject). If it is not Medical Monitor in advance of tor must promptly document the case in rd. Subsequently, the Investigator cal Monitor to explain any premature assignment (eg, accidental unblinding or us AE [SAE]). Procedures for eatment will be provided separately to edical Monitor will document within a rationale, circumstances, and the dabout the unblinding. |
| 9.7.1 Visit<br>Windows | (Week 1 Visit) to confirm eligibility. Subjects who have not taken statins within 4 weeks of Screening Visit 1 are not required to enter into the washout period and may proceed to Screening Visit 2 (Week 1) to provide a fasting blood sample. The Week 1 Visit should occur within ±1 days of the Randomization/Day1 | | Randomization/Day 1 V<br>the time of screening or required to stop statin the provide a fasting blood s eligibility. Subjects who of Screening Visit 1 are period and may proceed blood sample. The Randomization of Screening Visit 1 are period and may proceed blood sample. | nts should occur ≤35 days prior to the Visit. Subjects who are taking statins at within 30 days of Screening Visit 1 are crapy for 4 weeks (28 (±1) days), and ample at Screening Visit 2 to confirm have not taken statins within 30 days not required to enter into the washout to Screening Visit 2 to provide a fasting lomization/Day 1 Visit may occur as os are available and eligibility is |
| | Visit or Procedure | Visit Window and/or Interval | X/: -:4 D d | V'-'4 W'-11 |
| | Screening Visit 1 | Visit(s) are to occur ≤5 weeks (35 days) before Day 1. | Screening Visit 1 | Visit Window and/or Interval Visit(s) are to occur ≤5 weeks |
| | LTSE Visits: Month 3,<br>Month 6, Month 9,<br>Month 12, Month 15,<br>Month 18, and<br>Month 21 | ±1 week (7 days); the LTSE visits are relative to LTSE Day 1 (ie, Week 16 of double-blind phase) | Screening visit 1 | (35 days) <b>prior</b> to Day 1. |

| Section | Original Text | Revised Text |
|---|---|---|
| | | LTSE Visits: Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, and Month 21 ±1 week (7 days); the LTSE visits are relative to LTSE Day 1 (ie, Week 16 of double-blind phase) |
| 9.7.3 Screening Visit 1 Procedures (≤35 Days Before Day 1) | The Screening Visit assessments must be performed within ≤5 weeks prior to Day 1 to determine whether the subject meets all the inclusion criteria and none of the exclusion criteria. Subjects who do not fulfill all eligibility criteria will not be enrolled in the study. | The Screening Visit assessments must be performed ≤5 weeks prior to Day 1 to determine whether the subject meets all the inclusion criteria and none of the exclusion criteria. Subjects who do not fulfill all eligibility criteria will not be enrolled in the study. |
| | Subjects who are statin-free (ie, no statin use within 4 weeks of Screening) must return for fasted serum chemistry labs at Screening Visit 2, and may proceed to the Randomization/Day 1 Visit once screening labs are available and eligibility is confirmed; subjects who need to wash out statin therapy are required to "have a Week -1 Visit 4 weeks after Screening Visit 1." Additional Screening Visit 1 procedure for subjects currently taking statins: • Subjects who are currently taking statins, defined as statin use within 4 weeks of Screening, will be instructed to discontinue statin therapy following Screening Visit 1. These subjects must complete a 5 week statin washout prior to being randomized. After 4 weeks of statin washout, subjects will return for Screening Visit 2/Week —1 Visit to provide blood samples for fasted serum chemistry. | Subjects who are statin-free (ie, no statin use within 30 days of Screening) must return for fasted serum chemistry labs at Screening Visit 2, and may proceed to the Randomization/Day 1 Visit once screening labs are available and eligibility is confirmed; subjects who need to wash out statin therapy are required to return for Screening Visit 2 following the washout period. Additional Screening Visit 1 procedure for subjects currently taking statins: • Subjects who are currently taking statins, defined as statin use within 30 days of Screening, will be instructed to discontinue statin therapy following Screening Visit 1. After 4 weeks of statin washout, subjects will return for Screening Visit 2 to provide blood samples for fasted serum chemistry. |
| 9.7.4 Screening<br>Visit 2 <del>/Week 1</del><br>Visit-Procedures | Subjects who were receiving statin therapy at the time of screening. • Verify that subjects have completed a 4-week washout period. | All subjects will return for Screening Visit 2 to confirm eligibility criteria and provide blood samples for fasted serum chemistry. For subjects who were receiving statin therapy at the time of |
| | All Subjects: | <ul> <li>Verify that subjects have completed a 4-week washout period.</li> </ul> |

| Section | Original Text | Revised Text |
|---|---|---|
| | | For all subjects: |
| 9.7.14 Additional<br>Procedures at<br>Week 16/LTSE | Subject who will continue into the LTSE phase after completing the procedures listed for the Week 16 Visit | Subjects who continue into the LTSE phase after completing the procedures listed for the Week 16 Visit |
| Day 1 | Dispense investigational product as instructed | <ul> <li>Record the visit in IWRS, randomize the subject to one<br/>of the open-label treatment groups, and dispense open-<br/>label investigational product according to IWRS<br/>instructions.</li> </ul> |
| 9.7.16 LTSE<br>Visits | LTSE Visits will occur every 3 months (eg, at Months 3, 6, 9, and 12) following completion of the Week 16/LTSE Day 1 Visit. The visit procedures described below will repeat annually for the duration of the LTSE. For example, once a subject completes a year (Month 12 Visit) in the LTSE, their next visit should be 3 months later and the procedures described for the Month 3 LTSE Visit should be followed. | LTSE Visits should occur within ±1 week of the visit day and the timing of all visits should be relative to the double-blind Week 16 Visit (ie, the start of the LTSE; LTSE Day 1). For example, if the Month 6 Visit occurred 1 week late, the Month 9 Visit should still be approximately 9 months after the Week 16 Visit. |
| 9.7.16 LTSE<br>Visits | LTSE Visits should occur within ±1 week of the visit day and the timing of all visits should be relative to the double blind Week 16 Visit (ie, the start of the LTSE; LTSE Day 1). For example, if the Month 6 Visit occurred 1 week late, the Month 9 Visit should still be approximately 9 months after the Week 16 Visit. | The first LTSE visit following LTSE Day 1 will occur at LTSE Month 1. The next visit will occur at LTSE Month 3 and every 3 months thereafter (eg, at Months 6, 9, and 12) for the duration of the LTSE. The quarterly visit procedures described below will repeat annually for the duration of the LTSE. For example, once a subject completes a year (Month 12 Visit) in the LTSE, their next visit should be 3 months later and the procedures described for the Month 3 LTSE Visit should be followed. |
| 9.7.17 LTSE<br>Month 1<br>Contact/Visit<br>Procedures | Approximately 1 month into the LTSE, the subject should be contacted to assess compliance with OCA treatment, review and record concomitant medications, and assess and record AEs. This is not a clinic visit. This contact is not repeated in subsequent years of participation. | <ul> <li>Verify that the subject has fasted for at least 8 hours.</li> <li>Record fasting status in the source and eCRF.</li> <li>If the subject reports having eaten within 8 hours, document accordingly in the source and eCRF and remind the subject that fasting is</li> </ul> |

| Section | Original Text | Revised Text |
|---|---|---|
| | | required prior to all study visits, but water is permitted. |
| | | <ul> <li>Assess and record vital signs (body temperature,<br/>sitting heart rate, respiratory rate, and sitting blood<br/>pressure).</li> </ul> |
| | | Assess and record AEs. |
| | | Review and record concomitant medications. |
| | | <ul> <li>Collect used bottles of investigational product, assess<br/>investigational product compliance, and perform<br/>investigational product accountability. Following<br/>product accountability, redispense the same bottle of<br/>investigational product for use until the next visit.</li> </ul> |
| | | Collect used bottles of atorvastatin, assess atorvastatin compliance, and perform atorvastatin accountability. Following atorvastatin accountability, if the subjects is continuing with the same dose of atorvastatin, redispense the same bottle for use until the next visit. |
| | | • NOTE: If atorvastatin dose is up-titrated or re-<br>initiated after dose interruption, a telephone safety<br>contact must be conducted 2 weeks following the<br>change in dose to assess for AEs, concomitant<br>medications, and investigational product and<br>atorvastatin compliance. |
| | | Obtain blood samples for: |
| | | <ul> <li>Serum chemistry (will include basic lipid panel and<br/>liver biochemistry panel), hematology, and<br/>coagulation</li> </ul> |
| | | Markers of glucose metabolism |
| | | • CPK, if myopathy suspected |

| Section | Original Text | Revised Text |
|---|---|---|
| | | <ul> <li>Perform a urine based β-hCG pregnancy test in<br/>female subjects of childbearing potential. Perform<br/>serum pregnancy test in females of childbearing<br/>potential if urine β-hCG pregnancy test is positive.</li> </ul> |
| | | <ul> <li>Reiterate dosing instructions for investigational product and advise the subject:</li> </ul> |
| | | Take the investigational product at approximately the same time each day |
| | | <ul> <li>NOT to take investigational product or<br/>atorvastatin (if applicable) or on the morning<br/>of the next visit</li> </ul> |
| | | <ul> <li>To bring the investigational product and<br/>atorvastatin (if applicable) bottle(s); s/he will<br/>dose at the clinic</li> </ul> |
| | | <ul> <li>To fast overnight (at least 8 hours) prior to the<br/>next visit. Fasting is required prior to all study<br/>visits, but water is permitted.</li> </ul> |
| 10<br>Study Medication<br>Materials and<br>Management | STUDY MEDICATION MATERIALS AND MANAGEMENT | INVESTIGATIONAL PRODUCT AND STUDY MEDICATION |
| 10.1<br>Investigational<br>Product (OCA or | 5 mg, 10-mg and 25-mg OCA tablets for the LTSE Phase will be supplied as white or yellow tablets. | 10-mg and 25-mg OCA tablets for the LTSE Phase will be supplied as white or yellow tablets. |
| Placebo) LTSE<br>Phase: | • White OCA tablets are round and debossed with "INT" on one side and "3547" on the other side. | • White OCA tablets are round and debossed with "INT" on one side and "3547" on the other side. |
| | •—5 mg yellow tablets: Round and debossed with "INT" on one side and "5" on the other side. | |

Version 4: 19 Dec 2016

| Section | Original Text | Revised Text | | | | |
|---|---|---|---|---|---|---|
| | <ul> <li>10 mg yellow tablets: Triangular and debossed with "INT" on one side and "10" on the other side.</li> <li>5 mg yellow tablets: Oval and debossed with "INT" on one side and "25" on the other side.</li> </ul> | | | | | |
| 10.3<br>Investigational<br>Product Storage | Investigational product should be stored at the clinical study sites in the containers in which they are received from the Sponsor's supplier, at 15-25°C and protected from excess humidity. | Investigational product should be stored in the containers in which they are received from the Sponsor's supplier, at 15-2 | | | | |
| 11.1.2.1 Central<br>Reading of Liver<br>Histology | All biopsy assessments, including determination of study eligibility based on NASH diagnosis and fibrosis staging during Screening, will be performed centrally by an independent pathologist. Key features of NASH (ie, steatosis, lobular inflammation, and hepatocellular ballooning) will be graded in accordance with the NASH CRN criteria for scoring (Kleiner 2005). Fibrosis staging for eligibility will also be performed in accordance with NASH CRN criteria for fibrosis staging. | Screening, will be performed centrally by an independent pathologist. <b>The central pathologist must confirm</b> | | | osis staging during independent onfirm num NAS of 4 t of NAS. Key mmation, and ccordance with the 5) as summarized ll also be | |
| | | NAFLD Activity Score (NAS) Fibrosis Sta | | osis Staging | | |
| | | | Parameter | Scoring<br>Criteria | Paramete<br>r | Staging<br>Criteria |

| Original Text | | | | |
|---|---|---|---|---|
| | Steatosis | 0 = <5%<br>1 = 5% -<br>33%<br>2 = >33%<br>- 66%<br>3 = >66% | Stage 0 | No Fibrosis |
| | Lobular<br>Inflammatio<br>n | 0 = No Foci 1 = <2 Foci per 200 × field 2 = 2-4 Foci per 200 × field 3 = > 4 Foci per 200 × field | Stage 1<br>Stage 1a<br>Stage 1b<br>Stage 1c | Perisinusoidal or Periportal Mild, zone 3, persinusoidal Moderate, zone 3, perisinusoida l Portal / periportal |
| | Ballooning | 0 = None<br>1 = Few<br>balloon | Stage 2 | Perisinusoidal<br>and portal /<br>periportal |
| | | cells 2 = Many | Stage 3 | Bridging<br>fibrosis |
| | | cells / prominen t balloonin | Stage 4 | Cirrhosis |
| _ | Original Text | Lobular Inflammatio n | Steatosis | Steatosis |

Version 4: 19 Dec 2016

| Section | Original Text | Revised Text |
|---|---|---|
| | | scoring (Ishak 1995) for all subjects. Any extra biopsy tissue may undergo exploratory histological evaluations. |
| 11.2.2<br>Pharmacokinetic<br>Assessments | The first sample should be collected within 30 minutes prior to administration of investigational product (predose) on Day 1 at the Week 16 Visit. | The first sample should be collected within 30 minutes prior to administration of investigational product (predose) on Day 1 and prior to administration of investigational product or atorvastatin at the Week 16 Visit. |
| 12.1.2<br>Relationship to<br>Investigational<br>Product or Study<br>Medication | | If the relationship between a SAE and the atorvastatin is determined to be "definite," "probable," or "possible," the event will be considered to be related to atorvastatin for the purpose of assessing expedited safety reporting and reporting to the manufacturer. |
| 12.1.4.1 Severity<br>of Pruritus (as<br>and AE) | | Since pruritus is a subjective symptom and the occurrence and magnitude of which are not readily measured by objective tools, clinical judgment needs to be applied in the management of each subject. Managing OCA-related pruritus may help improve tolerance in those subjects who experience problematic pruritus and may otherwise discontinue from the study prematurely. General guidance for the management of subjects experiencing significant pruritus includes: |
| | | Drug holiday: A drug holiday is defined as an Investigator 'prescribed' complete interruption of dosing for 1 or more consecutive days (ie, non-daily dosing does not constitute a drug holiday). For subjects with severe pruritus, instruct the subject to stop taking investigational product until the pruritus subsides to an acceptable level, at which time it should be restarted. Details of drug holidays and/or nondaily dosing regimens should be recorded in the CRF. |
| | | Prescribe BAS. Subjects taking BAS (including colestyramine and its derivatives, colestipol, colesevelam, or other sequestrants) should be |

| Section | Original Text | Revised Text |
|---|---|---|
| | | <ul> <li>instructed to stagger their dosing of investigational product, ensuring at least 4 hours between doses of the BAS and investigational product.</li> <li>Other therapies may be tried as deemed clinically</li> </ul> |
| | | appropriate. |
| | | <ul> <li>Less frequent dosing of investigational product (eg,<br/>on alternate days) may be tried, after which subjects<br/>may return to their original daily dose as soon as<br/>tolerated.</li> </ul> |
| 12.1.8.1<br>Pregnancy and<br>Follow-Up | Pregnancies are not considered AEs in and of themselves; however, if a female study participant becomes pregnant while she is enrolled in the clinical study, she must discontinue treatment with investigational product and atorvastatin immediately (see Section 8.4.1.1) and the Sponsor must be notified within 24 hours of the Investigator's learning of the pregnancy by completing the Pregnancy Report eCRF in the EDC system.—Entering the pregnancy report into the EDC system will automatically notify the Sponsor of the pregnancy.—The subject and neonate must be followed for outcome information and/or as considered appropriate by the Investigator and the Sponsor. Women who discontinue the study due to pregnancy may not reenroll in the study at any point, but should continue with the study visit schedule and must be followed by the Investigator through pregnancy outcome. Similarly, if a subject's pregnancy is terminated early (planned or unplanned), the subject will also be removed from the study. Completing the Pregnancy Report in the EDC is not a substitute for reporting an AE/SAE when an AE/SAE has occurred. In the situation when an AE/SAE has occurred, the AE/SAE reporting procedures described in Section 17.1 must also be followed. | Pregnancies are not considered AEs in and of themselves; however, if a female study participant becomes pregnant while she is enrolled in the clinical study, she must discontinue treatment with investigational product and atorvastatin immediately (see Section 8.4.1.1) and the Sponsor must be notified within 24 hours of the Investigator's awareness of the pregnancy by completing the Pregnancy eCRF in the EDC system and downloading and completing the Pregnancy Report Form. The Pregnancy Report Form must be emailed to sae@interceptpharma.com or faxed to +1-800-497-8521. The subject and neonate must be followed for outcome information and/or as considered appropriate by the Investigator and the Sponsor. Women who discontinue the study due to pregnancy may not reenroll in the study at any point, but should continue with the study visit schedule and must be followed by the Investigator through pregnancy outcome. Similarly, if a subject's pregnancy is terminated early (planned or unplanned), the subject will also be removed from the study. Completing the Pregnancy Report Form is not a substitute for reporting an AE/SAE if an AE/SAE has occurred related to or concurrent with the pregnancy. In the situation when an AE/SAE has occurred, the AE/SAE reporting procedures described in Section 1.7.1 must also be followed. |

| Section | Original Text | Revised Text |
|---|---|---|
| 12.2.4<br>Electrocardiogra<br>m | Investigative sites must retain a copy of all 12-lead ECGs evaluated by the Investigator or designee. These ECGs must be clearly labeled with the subject's initials, Subject ID number, date, and time. Full instructions will be provided for forwarding the 12-lead ECGs for central reading. | Investigative sites must retain a copy of all 12-lead ECGs evaluated by the Investigator or designee. These ECGs must be clearly labeled with the Subject ID number, date, and time. Full instructions will be provided for forwarding the 12-lead ECGs for central reading. |
| 12.2.6 Laboratory<br>Assessments | Except for Screening, subjects will be instructed to attend each study visit in a fasted state, and subjects should remain fasted until their blood samples have been collected. | Except for Screening <b>Visit 1</b> , subjects will be instructed to attend each study visit in a fasted state, and subjects should remain fasted until their blood samples have been collected. |
| 13.6.3.7<br>Pharmacokinetic<br>Analysis | The PK Population will be used for analysis of PK parameters, which include plasma OCA (parent) and its conjugates (glyco-OCA and tauro-OCA), total OCA, and potentially other conjugates or metabolites not yet identified. PK analysis will be done using non-compartmental methods. | The PK Population will be used for analysis of PK parameters, which include plasma OCA (parent) and its conjugates (glyco-OCA and tauro-OCA), total OCA, <b>OCA glucuronide</b> and potentially other conjugates or metabolites not yet identified. PK analysis will be done using non-compartmental methods. |
| 13.7.5<br>Adjudicated<br>Cardiovascular<br>Events | | Adjudicated cardiovascular events include core MACE (cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke) and expanded MACE (unstable angina requiring hospitalization, transient ischemic attack, peripheral or coronary revascularization procedures, hospitalization for congestive heart failure). Other events potentially related to adverse cardiovascular outcomes are defined in Appendix D and will be included in the Cardiovascular Adjudication Committee Charter for adjudication. Undetermined cause of death will be classified as a cardiovascular death by the Cardiovascular Adjudication Committee. |
| | | Summaries of adjudicated cardiovascular events will include the incidence of TEAEs and the incidence of serious TEAEs. All summaries of incidence will include the associated exact binomial 95% CI. |
| 13.9 Adjudication<br>Committees | Cardiovascular Events-Committee (CEC): Adjudicates all suspected MACE | Cardiovascular Adjudication Committee (CAC): Adjudicates all suspected MACE, including all deaths |
| 16.4 Subject<br>Confidentiality | All information obtained during the conduct of the study with respect to the subject will be regarded as confidential and | All information obtained during the conduct of the study with respect to the subject will be regarded as confidential and |

| Section | Original Text | Revised Text |
|---|---|---|
| and Data<br>Protection | confidentiality of all subjects will be maintained. Monitors (eg, CRA, Medical Monitor), auditors and inspectors will require access to a subject's medical notes for the purpose of source document verification but the subject's confidentiality will be maintained at all times. An agreement for disclosure of any such information will be obtained in writing and is included in the statement of informed consent. The study data shall not be disclosed to a third party (with the exception of auditors and/or regulatory authorities) without the written consent of the Sponsor. All data shall be secured against unauthorized access. The Investigator will maintain a list of subject names and identifying information (eg, subjects' hospital numbers, unique subject numbers). This list will not be collected by the Sponsor. The written information sheet will explain that study data will be stored in a computer database, maintaining confidentiality in accordance with national data protection legislation. All data computer processed by the Sponsor or designee will be identified by unique subject number/randomization code/subject initials/site number, only. | confidentiality of all subjects will be maintained. Monitors (eg, CRA, Medical Monitor), auditors and inspectors will require access to a subject's medical notes for the purpose of source document verification but the subject's confidentiality will be maintained at all times. An agreement for disclosure of any such information will be obtained in writing and is included in the statement of informed consent. The study data shall not be disclosed to a third party (with the exception of auditors and/or regulatory authorities) without the written consent of the Sponsor. All reports and communications relating to subjects in this study that are disclosed to an authorized third party will identify subjects only by protocol and assigned number and will be shared in a secure manner. All data shall be secured against unauthorized access. The Investigator will maintain a list of subject names and identifying information (eg, subjects' hospital numbers, unique subject numbers). This list will not be collected by the Sponsor. The written information sheet will explain that study data will be stored in a computer database, maintaining confidentiality in accordance with national data protection legislation. All data computer processed by the Sponsor or designee will be identified by unique subject number/randomization code/ site number, only. |
| 19 List of<br>References | | Beuers U, Gershwin ME, Gish RG, et al. Changing nomenclature for PBC: From 'cirrhosis' to 'cholangitis'. Dig Liver Dis. 2015a;47(11):924-6. Beuers U, Gershwin ME, Gish RG, et al. Changing nomenclature for PBC: From 'cirrhosis' to 'cholangitis'. Gastroenterology. 2015b;149(6):1627-9. |
| | | Beuers U, Gershwin ME, Gish RG, et al. Changing nomenclature for PBC: From 'cirrhosis' to 'cholangitis'. Hepatology. 2015c;62(5):1620-2. |

| Section | Original Text | Revised Text |
|---|---|---|
| Appendix D | Appendix D included Major Adverse Cardiovascular Event Definitions from Chapters 1 through 7 of "Standardized Definitions for Cardiovascular and Stroke Endpoint Events in Clinical Trials," dated August 20, 2014 | Appendix D was updated to add definitions from Chapters 8 through 10 of "Standardized Definitions for Cardiovascular and Stroke Endpoint Events in Clinical Trials," dated August 20, 2014 |

## APPENDIX H. 747-209 PROTOCOL VERSION 4 SUMMARY OF CHANGES

Protocol 747-209 was revised to include the following information:

- Incorporation of the evaluation the bioanalytical concentrations of atorvastatin and its metabolites.
- Updating the maximum percentage of subjects with stage 4 fibrosis from 20% to 30%.
- Removing the obeticholic acid (OCA) glucuronide component of PK as that bioanalysis will be conducted in another study.
- Additional clarifications.

## **Summary of Changes**

The following revisions were made to the protocol in Protocol Version 4. Revised and new text in Version 4 is indicated in **bold** font, and the text deleted from Protocol Version 3 is crossed out in the table below. Minor/editorial changes are not listed individually in the summary table below.

| Section | Original Text (Version 3) | Revised Text (Version 4) | Key Change<br>Reasons /<br>Justification for Change |
|---|---|---|---|
| Study Personnel<br>Contact Information | Investigators are encouraged to call the NASH medical monitor hotline at +1 844 250 6396 or send an email to the NASH medical monitor at NASH209@interceptpharma.com with safety questions as these lines of contact are monitored 24 hours a day. The following individual medical monitors may also be contacted through the NASH medical monitor hotline and email address. | Investigators are encouraged to call the PRA Medical Support Center phone number for the United States and Canada at +1 866 326 5053 or send an email to the NASH medical monitor at CONTROL@prahs.com with safety questions as these lines of contact are monitored 24 hours a day. | The PRA Medical Support<br>Center phone number and<br>email address were updated. |

| Section | Original Text ( | Version 3) | Revised Text (Ver | rsion 4) | Key Change<br>Reasons /<br>Justification for Change |
|---|---|---|---|---|---|
| Study Personnel<br>Contact Information | NASH<br>Medical<br>Monitor<br>Hotline<br>Email | +1 844 250 6396 NASH209@interceptpharma.com | Deletion | | Removed the NASH Medical<br>Monitor Hotline Email (no<br>longer applicable). |
| Study Personnel<br>Contact Information | Primary Medical Monitor Contact: Phone: Email Secondary Contact: Mobile Phone: Email | Emad Basta, MD (Lead) Medical Monitor/Medical Expert PRA Health Sciences +1 866 326 5053 CONTROL@PRAHS.com Roya Hooshmand Rad, MD PhD Executive Director, Medical Safety and Pharmacovigilance Intercept Pharmaceuticals, Inc. (Intercept) +1 858 880 6485 (Pacific time zone) rhooshmand rad @interceptpharma.com | Primary Medical<br>Monitor Contact: Phone: Email Secondary Contact: Mobile Phone: Email | Emad Basta, MD (Lead) Medical Monitor/Medical Expert PRA Health Sciences +1 866 326 5053 CONTROL@prahs.com Tolga Baykal, MD, PhD Medical Director, Clinical Development Intercept Pharmaceuticals, Inc. (Intercept) +1 619 643 8886 (Pacific time zone) tolga.baykal@interceptpharma.c om | Updated email address. Tolga Baykal was added as secondary contact. |
| Synopsis Objectives: Exploratory Objectives 6.3 Exploratory Objectives | Insertion | | To evaluate the bioanalytical concentrations of atorvastatin and its metabolites | | New exploratory objective for<br>the determinations of the<br>concentrations of atorvastatin<br>and its metabolites. |
| Synopsis<br>Number of Subjects<br>(Planned) | NASH and evid<br>decompensation<br>randomized in a | 80 subjects with biopsy-confirmed ence of liver fibrosis, but no hepatic, who meet eligibility criteria, will be 1:1:1:1 ratio to 1 of 4 treatment mum of 20% of subjects will have | Approximately 80 subjects with biopsy-confirmed NASH and evidence of liver fibrosis, but no hepatic decompensation, who meet eligibility criteria, will be randomized in a 1:1:1:1 ratio to 1 of 4 treatment groups. A maximum of 30% of subjects will have stage 4 fibrosis. | | The rapid rate of enrollment of subjects with stage 4 fibrosis allowed patients already in screening to be enrolled after the initial maximum of 20% was met (the overall number of subjects remains at $\sim$ 80). |

| Section | Original Text (Ver | sion 3) | Revised Text (Version 4) | | Key Change<br>Reasons /<br>Justification for Change |
|---|---|---|---|---|---|
| Synopsis<br>Statistical Methods<br>11.1, Efficacy<br>Assessments | OCA pharmacokinetics | OCA, tauro-OCA, glyco-OCA, total OCA <del>, OCA glucuronide</del> , potentially other conjugates or metabolites not yet identified | OCA pharmacokinetics | OCA, tauro-OCA, glyco-OCA, total OCA, potentially other conjugates or metabolites not yet identified | Removal of OCA glucuronide as that bioanalysis will be conducted in another study. |
| Table 4, List of Planned Assessments | Insertion | | Exploratory Endpo | ints | Addition of the determination |
| | | | Atorvastatin<br>bioanalytical<br>concentrations | Atorvastatin and its metabolites | of the concentration of atorvastatin and its metabolites to characterize atorvastatin concentrations with and without OCA. |
| Synopsis<br>Analysis Populations<br>13.1, Analysis Sets | consent to participat<br>at least one confirm<br>Subjects must have<br>hours before the vis | pulation: will include all OCA subjects who te in the PK assessments and have ed fasted analyzable sample. been fasting for approximately 8 it and must not have any major that potentially affect exposure | Pharmacokinetic Populations: The OCA PK Population will include all OCA subjects who consent to participate in the PK assessments and have at least one confirmed fasted analyzable sample. Subjects must have been fasting for approximately 8 hours before the visit and must not have any major protocol deviations that potentially affect exposure levels. The Atorvastatin PK Population will include all subjects who consent to participate in the PK assessments and have at least one confirmed fasted analyzable sample. | | Differentiation of OCA PK<br>Population and incorporation<br>of the Atorvastatin PK<br>Population. |
| 7.1.2, Schedule of<br>Study Procedures<br>Table 1, Schedule of<br>Study Procedures:<br>Double-Blind Period | option to provide blooms PK. PK samp minutes prior to dos 2.5, 3, 4, 5, and 6 he drink additional wat | gational sites, subjects will have the ood samples for measurement of les will be collected within 30 ing and again at 0.5, 0.75, 1, 1.5, 2, ours postdose. Subjects should not ter for 1 hour after taking the dose oduct and will remain fasted until a collected. | s At selected investigational sites, subjects will have the option to provide blood samples for measurement of PK for OCA (Day 1 and Week 16), and for atorvastatin (Week 16). PK samples will be collected within 30 minutes prior to dosing and again at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. Subjects should not drink additional water for 1 hour after taking the dose of investigational product and will remain fasted until the 1 hour sample is collected. | | Clarification on the PK sampling of OCA and incorporation of atorvastatin PK sampling. |
| 7.2, Number of Subjects | criteria, including be<br>evidence of liver fib<br>decompensation, wi | ubjects who meet the eligibility iopsy-confirmed NASH and prosis, but no hepatic ll be included in this study. A f subjects will have stage 4 fibrosis. | Approximately 80 subjects who meet the eligibility criteria, including biopsy-confirmed NASH and evidence of liver fibrosis, but no hepatic decompensation, will be included in this study. A maximum of 30% of subjects will have stage 4 fibrosis. | | The rapid rate of enrollment of subjects with stage 4 fibrosis allowed patients already in screening to be enrolled after the initial maximum of 20% |

| Section | Original Text (Version 3) | Revised Text (Version 4) | Key Change Reasons / Justification for Change was met (the overall number of subjects remains at ~ 80). |
|---|---|---|---|
| 9.7.13.1, Additional<br>Week 16 Procedures<br>for PK Subjects | Following collection of the Week 16 fasted samples indicated above, subjects who are participating in the PK assessment will each receive a single dose of their assigned investigational product with water. Serial blood samples will be obtained for measurement of OCA and its conjugates 30 minutes prior to dosing and at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. | Following collection of the Week 16 fasted samples indicated above, subjects who are participating in the PK assessment will each receive a single dose of their assigned <b>double-blind</b> investigational product with water. Serial blood samples will be obtained for measurement of OCA and its conjugates, <b>and atorvastatin and its metabolites</b> , 30 minutes prior to dosing and at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. | Clarification of study phase. Incorporation of PK sampling for atorvastatin. |
| 11.2,<br>Pharmacokinetic and<br>Pharmacodynamic<br>Assessments | Parent OCA and its major conjugates (glyco-OCA and tauro-OCA), C4, and FGF-19 concentrations will be determined for OCA PK and FXR activity in OCA-treated subjects. Samples will be obtained for possible assessment of conjugated and unconjugated bile acids. | Parent OCA and its major conjugates (glyco-OCA and tauro-OCA), C4, and FGF-19 concentrations will be determined for OCA PK and FXR activity in OCA-treated subjects. Concentrations of atorvastatin and its metabolites will be assessed in PK sampled subjects. Samples will be obtained for possible assessment of conjugated and unconjugated bile acids. | Addition of the determination of the concentration of atorvastatin and its metabolites. |
| 11.2.2,<br>Pharmacokinetic<br>Assessments | Subjects who opt to participate in the PK assessment will provide blood samples for the measurement of OCA and its conjugates. The first sample should be collected within 30 minutes prior to administration of investigational product (predose) on Day 1 and prior to administration of investigational product or atorvastatin at the Week 16 Visit. Subjects will then receive a single dose of investigational product with approximately 240 mL of water. Serial blood samples will be obtained for measurement of OCA and its conjugates at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. | Subjects who opt to participate in the PK assessment will provide blood samples for the measurement of OCA and its conjugates, and atorvastatin and its metabolites. The first sample should be collected within 30 minutes prior to administration of investigational product (predose) on Day 1 and prior to administration of investigational product or atorvastatin at the Week 16 Visit. Subjects will then receive a single dose of investigational product with approximately 240 mL of water. Serial blood samples will be obtained for measurement of OCA and its conjugates, and atorvastatin and its metabolites, at 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, and 6 hours postdose. | Incorporation of atorvastatin PK and sampling. |

| Section | Original Tex | t (Version 3) | Revised Text (Version 4) | | Key Change<br>Reasons /<br>Justification for Change |
|---|---|---|---|---|---|
| 12.1.4.1, Severity of Pruritus (as an AE) | •Drug holiday: A drug holiday is defined as an Investigator 'prescribed' complete interruption of dosing for 1 or more consecutive days (ie, non-daily dosing does not constitute a drug holiday). For subjects with severe pruritus, instruct the subject to stop taking investigational product until the pruritus subsides to an acceptable level, at which time it should be restarted. Details of drug holidays and/or nondaily dosing regimens should be recorded in the CRF. | | •Drug holiday: A drug holiday is defined as an Investigator 'prescribed' complete interruption of dosing for 1 or more consecutive days (ie, non-daily dosing does not constitute a drug holiday). Details of drug holidays and/or nondaily dosing regimens should be recorded in the CRF. Per Section 8.4.1.1, subjects with pruritus ≥Grade 3 in severity and possibly, probably, or definitely related to investigational product must discontinue investigational product. | | Instructions for severity of pruritus were removed. The instructions for the handling of ≥Grade 3 in severity are provided. |
| 12.2.6, Laboratory<br>Assessments<br>Table 10, List of<br>Laboratory Analytes | Subset of Subjects | | Subset of Subjects | | Removal of OCA glucuronide. |
| | PK analytes | OCA, tauro-OCA, glyco-OCA, OCA glucuronide and possible other conjugates or metabolites not yet | PK analytes | OCA, tauro-OCA, glyco-OCA,<br>and possible other conjugates or<br>metabolites not yet identified | Addition of atorvastatin and its metabolites. |
| to be Tested | | identified | | Atorvastatin and its metabolites | |
| | VLDL choles<br>particle conc<br>ApoCII, Apo<br>chemistry pa | panel will be used for (a) LDL, HDL, and sterol concentrations, particle sizes, and entrations, and (b) ApoA1, ApoB, ApoE, CIII and Lp(a) concentrations. Serum nel will be used for LDL, HDL, VLDL, I cholesterol concentration. | <sup>a</sup> NMR-based panel will be used for LDL, HDL, and VLDL cholesterol concentrations, particle sizes, and particle concentrations. ApoA1, ApoB, ApoE, ApoCII, ApoCIII, Lp(a) and PCSK9 concentrations will be measured using appropriate methods at central or specialty laboratories. Serum chemistry panel will be used for LDL, HDL, VLDL, TG, and total cholesterol concentration. | | Clarification of methods to be used for the determination of ApoA1, ApoB, ApoE, ApoCII, ApoCIII, Lp(a), and PCSK9 concentrations. |
| 13.6.3.7,<br>Pharmacokinetic<br>Analysis | parameters, with conjugates (gloch glucuror metabolites not using non-con The values with group using do have a confirm more before the Further details | ation will be used for analysis of PK hich include plasma OCA (parent) and its yco-OCA and tauro-OCA), total OCA, nide, and potentially other conjugates or by yet identified. PK analysis will be done inpartmental methods. Il be summarized by active treatment escriptive statistics. Only samples that need fasting of approximately 8 hours or neir visit will be included in the analysis. It regarding specific parameters and the described in the SAP. | The PK Population will be used for analysis of PK parameters, which include plasma OCA (parent) and its conjugates (glyco-OCA and tauro-OCA), total OCA, atorvastatin and its metabolites, and potentially other analytes not yet identified. PK analysis will be conducted using standard non-compartmental methodologies. For the analysis of OCA and its conjugates, values will be summarized by active treatment group using descriptive statistics. Only samples that have a confirmed fasting of approximately 8 hours or more before their visit will be included in the analysis. | | Incorporation of clarifications for OCA and atorvastatin PK analysis. |

| Section | Original Text (Version 3) | Revised Text (Version 4) | Key Change<br>Reasons /<br>Justification for Change |
|---|---|---|---|
| | | Further details regarding the methods for calculating PK and the specific parameters to be reported will be described in the SAP. | |